Official Title: Phase I Study of the Combination of Trastuzumab Emtansine (T-

DM1) and Capecitabine in HER2-Positive Metastatic Breast Cancer and HER2-Positive Locally Advanced/Metastatic Gastric Cancer Patients, Followed by a Randomized, Open-Label Phase II Study of Trastuzumab Emtansine and Capecitabine Versus Trastuzumab Emtansine Alone in HER2-Positive Metastatic

**Breast Cancer** 

NCT Number: NCT01702558

**Document Dates:** Protocol Amendment Version 4: 23-Mar-2016

Protocol Amendment Version 3: 30-Jun-2014

Protocol Amendment Version 2: 03-Sep-2013

Protocol Version 1: 02-Jul-2012

# 13.1.1 Protocol and Protocol Amendments

The following documents are included in this appendix:

| Protocol | Version 1 | 02 Jul 2012 |
|------------------------------|---------------|-------------|
| Protocol | Version 2 | 03 Sep 2013 |
| Note to File for Version 2 | Note to File | 22 Oct 2013 |
| Protocol | Version 3 | 30 Jun 2014 |
| Protocol | Version 4 | 23 Mar 2016 |
| Protocol Amendment Version 2 | Final Version | 03 Sep 2013 |
| Protocol Amendment Version 3 | Final Version | 30 Jun 2014 |
| Protocol Amendment Version 4 | Final Version | 23 Mar 2016 |

#### PROTOCOL

TITLE: PHASE I FOLLOWED BY PHASE II STUDY OF THE COMBINATION

OF TRASTUZUMAB EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED OR METASTATIC GASTRIC

**CANCER PATIENTS** 

PROTOCOL NUMBER: MO28230 VERSION NUMBER: 1

**EUDRACT NUMBER:** 2012-001547-46

TEST PRODUCT: Trastuzumab emtansine (RO5304020)

MEDICAL MONITOR: MD

SPONSOR: F. Hoffmann-La Roche Ltd

DATE FINAL: See electronic date stamp below

### FINAL PROTOCOL APPROVAL




The information contained in this document, especially any unpublished data, is the property of F. Hoffmann-La Roche Ltd (or under its control) and therefore is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Ethics Committee or Institutional Review Board. It is understood that this information will not be disclosed to others without written authorization from Roche except to the extent necessary to obtain informed consent from persons to whom the drug may be administered.

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 1

# **TABLE OF CONTENTS**

| PR | OTOCOL AC | CCEPTANCE FORM | 9 |
|---|---|---|---|
| PR | OTOCOL SY | NOPSIS | 10 |
| 1. | BACKGRO | UND | 24 |
| | 1.1 | Background on Disease | 24 |
| | 1.1.1 | HER2-Positive Breast Cancer, Metastatic Breast Cancer | 24 |
| | 1.1.2 | HER2-Positive Locally Advanced or Metastatic Gastric Cancer | 25 |
| | 1.2 | Background on Study Drugs | 26 |
| | 1.2.1 | Trastuzumab Emtansine | 26 |
| | 1.2.1.1 | Study TDM3569g | 28 |
| | 1.2.1.2 | Study TDM4258g | 28 |
| | 1.2.1.3 | Study TDM4374g | 29 |
| | 1.2.1.4 | Study TDM4450g | 30 |
| | 1.2.1.5 | Study TDM4688g | 30 |
| | 1.2.1.6 | Phase III Study TDM4370g | 31 |
| | 1.2.1.7 | Pharmacokinetics | 32 |
| | 1.2.2 | Capecitabine | 34 |
| | 1.2.2.1 | Study BO18255: Capecitabine and Trastuzumab in mGC | 34 |
| | 1.2.3 | Preclinical Data of the Combination of Trastuzumab Emtansine and a Fluoropyrimidine | 35 |
| | 1.3 | Study Rationale and Benefit-Risk Assessment | |
| | 1.3.1 | For mBC | 37 |
| | 1.3.2 | For mGC | 38 |
| 2. | OBJECTIV | ES | 39 |
| | 2.1 | Phase I: MTD Finding of Trastzumab Emtansine and Capecitabine in mBC | 39 |
| | 2.1.1 | Primary Objective | 39 |
| | 2.1.2 | Secondary Objectives | |
| | 2.2 | Phase II: Exploration of Efficacy in mBC Patients | |
| | 2.2.1 | Primary Objective | 39 |
| | 2.2.2 | Secondary Objectives | 39 |

| | 2.3 | Phase I: MTD Finding of Trastzumab Emtansine and Capecitabine in MGC | 39 |
|---|---|---|---|
| | 2.3.1 | Primary Objective | |
| | 2.3.2 | Secondary Objectives | |
| 3. | STUDY DES | IGN | |
| | 3.1 | Description of Study | 40 |
| | 3.1.1 | Overview of Study Design | 40 |
| | 3.1.1.1 | Overview of Phase I Design in mBC Patients | 43 |
| | 3.1.1.2 | Overview of Phase II: Exploration of Efficacy in mBC Patients | 45 |
| | 3.1.1.3 | Overview of Phase I Design in mGC Patients | 45 |
| | 3.1.1.4 | Considerations for all Patients Treated in the Study | 46 |
| | 3.1.1.5 | Number of Patients | 46 |
| | 3.1.1.6 | Number of Centers | 46 |
| | 3.1.2 | Steering Committee | 46 |
| | 3.2 | End of Study | 47 |
| | 3.3 | Rationale For Study Design | 47 |
| | 3.3.1 | Rationale for Patient Group Selection | 47 |
| | 3.3.1.1 | Rationale for Phase I | 47 |
| | 3.3.1.2 | Rationale for Phase II | 47 |
| | 3.3.2 | Rationale For Investigational Medicinal Dose Selection | 47 |
| | 3.3.2.1 | In mBC Patients | 47 |
| | 3.3.2.2 | In mGC Patients | 48 |
| | 3.3.2.3 | Rationale for Duration of Treatment | 48 |
| | 3.3.3 | Pharmacokinetic Sampling Rationale | 48 |
| | 3.4 | Outcome Measures | 49 |
| | 3.4.1 | Phase I: mBC | 49 |
| | 3.4.1.1 | Primary Efficacy Outcome Measure | 49 |
| | 3.4.1.2 | Secondary Efficacy Outcome Measure | 49 |
| | 3.4.1.3 | Primary Safety Outcome Measure | 49 |
| | 3.4.1.4 | Secondary Safety Outcome Measures | 49 |
| | 3.4.1.5 | Pharmacokinetic Outcome Measures | 49 |
| | 342 | Phase II: Exploration of Efficacy: mBC | 49 |

| | 3.4.2.1 | Primary Efficacy Outcome Measure | 49 |
|----|-----------|--------------------------------------------------|------|
| | 3.4.2.2 | Secondary Efficacy Outcome Measures | 50 |
| | 3.4.2.3 | Primary Safety Outcome Measure | 50 |
| | 3.4.2.4 | Secondary Safety Outcome Measures | 50 |
| | 3.4.2.5 | Pharmacokinetic Outcome Measures | 50 |
| | 3.4.3 | Phase I: mGC | 50 |
| | 3.4.3.1 | Primary Efficacy Outcome Measure | 50 |
| | 3.4.3.2 | Secondary Efficacy Outcome Measure | 51 |
| | 3.4.3.3 | Primary Safety Outcome Measure | 51 |
| | 3.4.3.4 | Secondary Safety Outcome Measures | 51 |
| | 3.4.3.5 | Pharmacokinetic Outcome Measures | 51 |
| 4. | MATERIALS | S AND METHODS | . 51 |
| | 4.1 | Patients | . 51 |
| | 4.1.1 | mBC Patients | . 51 |
| | 4.1.2 | mGC Patients | 52 |
| | 4.1.3 | Inclusion Criteria | . 52 |
| | 4.1.3.1 | For mBC Patients | 52 |
| | 4.1.3.2 | For mGC Patients: | 53 |
| | 4.1.4 | Exclusion Criteria | 54 |
| | 4.1.4.1 | For mBC Patients: | 54 |
| | 4.1.4.2 | For mGC Patients: | 56 |
| | 4.2 | Study Treatment | 58 |
| | 4.2.1 | Formulation, Packaging, and Handling | 58 |
| | 4.2.1.1 | Trastuzumab Emtansine | 58 |
| | 4.2.1.2 | Capecitabine | 59 |
| | 4.2.2 | Dosage and Administration | 59 |
| | 4.2.2.1 | For mBC Patients | 59 |
| | 4.2.2.2 | For mGC Patients | 60 |
| | 4.2.3 | Investigational Medicinal Product Accountability | . 60 |
| | 4.2.4 | Post-trial Access to Extension Study | 61 |
| | 4.3 | Concomitant And Excluded Therapies | 61 |
| | 4.3.1 | Permitted Therapy | 61 |
| | 4.3.2 | Prohibited Therapy | 61 |
| | 4.4 | Study Assessments | 62 |
| | 4.4.1 | Description of Study Assessments | 62 |

| | 4.4.1.1 | Medical History and Demographic Data | . 62 |
|---|---|---|---|
| | 4.4.1.2 | Vital Signs | . 63 |
| | 4.4.1.3 | Physical Examinations | . 63 |
| | 4.4.1.4 | Tumor and Response Evaluations | . 63 |
| | 4.4.1.5 | Laboratory Assessments | . 64 |
| | 4.4.1.6 | Electrocardiograms | . 64 |
| | 4.4.1.7 | ECHO/MUGA | . 65 |
| | 4.4.2 | Timing of Study Assessments | . 65 |
| | 4.4.2.1 | Screening and Pretreatment Assessments | . 65 |
| | 4.4.2.2 | Assessments During Treatment | . 65 |
| | 4.4.2.3 | Assessments at Study Completion/Early Termination Visit | . 66 |
| | 4.4.2.4 | Follow-Up Assessments | . 66 |
| | 4.4.2.5 | Assessments at Unplanned Visits | . 67 |
| | 4.5 | Patient, Study, and Site Discontinuation | . 67 |
| | 4.5.1 | Patient Discontinuation | . 67 |
| | 4.5.2 | Study Discontinuation | . 67 |
| 5. | ASSESSME | NT OF SAFETY | |
| | 5.1 | Safety Plan | . 68 |
| | 5.1.1 | Risks Associated with Trastuzumab Emtansine | 68 |
| | 5.1.2 | Risks Associated with Capecitabine | . 70 |
| | 5.1.3 | Trastuzumab Emtansine and Capecitabine Combination: | . 70 |
| | 5.1.4 | Definition of Dose Limiting Toxicity | . 70 |
| | 5.1.5 | Management of Specific Adverse Events | . 71 |
| | 5.1.5.1 | Trastuzumab Emtansine Dosage Modification | . 71 |
| | 5.1.5.2 | Capecitabine Dosage Modification | . 77 |
| | 5.2 | Safety Parameters and Definitions | . 77 |
| | 5.2.1 | Adverse Events | . 77 |
| | 5.2.2 | Serious Adverse Events (Immediately Reportable to the Sponsor) | . 78 |
| | 5.2.3 | Protocol-Defined Events of Special Interest/Non-Serious Expedited Adverse Events | 79 |
| | 5 2 4 | Pregnancy and Contraception | 79 |

6.

| 5.3 | Methods and Timing for Capturing and Assessing Safety Parameters | 81 |
|---|---|---|
| 5.3.1 | Adverse Event Reporting Period | 81 |
| 5.3.2 | Eliciting Adverse Event Information | |
| 5.3.3 | Assessment of Severity of Adverse Events | 82 |
| 5.3.4 | Assessment of Causality of Adverse Events | |
| 5.3.5 | Procedures for Recording Adverse Events | 84 |
| 5.3.5.1 | Diagnosis Versus Signs and Symptoms | 85 |
| 5.3.5.2 | Adverse Events Occurring Secondary to other Events | 85 |
| 5.3.5.3 | Persistent or Recurrent Adverse Events | 85 |
| 5.3.5.4 | Abnormal Laboratory Values | 85 |
| 5.3.5.5 | Deaths | 86 |
| 5.3.5.6 | Pre-Existing Medical Conditions | 86 |
| 5.3.5.7 | Lack of Efficacy or Clinical Worsening | 87 |
| 5.3.5.8 | Hospitalization or Prolonged Hospitalization | 87 |
| 5.4 | Immediate Reporting Requirements from Investigator to the Sponsor | 87 |
| 5.4.1 | Emergency Medical Contacts | 88 |
| 5.4.2 | Reporting Requirements for Serious Adverse Events and Non-Serious Adverse Events of Special Interest | 88 |
| 5.4.3 | Reporting Requirements for Pregnancies | |
| 5.4.3.1 | Pregnancies in Female Patients | |
| 5.4.3.2 | Pregnancies in Female Partners of Male Patients | |
| 5.4.3.3 | Abortions | 80 |
| 5.4.3.4 | / (DOI (10110 | 09 |
| 5.4.5.4 | Congenital Anomalies/Birth Defects | |
| 5.4.3.4 | | 89 |
| | Congenital Anomalies/Birth Defects | 89<br>89 |
| 5.5 | Congenital Anomalies/Birth Defects Follow-Up of Patients after Adverse Events | 89<br>89 |
| 5.5<br>5.5.1 | Congenital Anomalies/Birth Defects | |
| 5.5<br>5.5.1<br>5.5.2 | Congenital Anomalies/Birth Defects | 89<br>89<br>90<br>90 |
| 5.5<br>5.5.1<br>5.5.2<br>5.6<br>5.7 | Congenital Anomalies/Birth Defects Follow-Up of Patients after Adverse Events Investigator Follow-Up Sponsor Follow-Up Post-Study Adverse Events Expedited Reporting to Health Authorities, Investigators, Institutional Review Boards, and Ethics Committees | 89<br>89<br>90<br>90 |
| 5.5<br>5.5.1<br>5.5.2<br>5.6<br>5.7 | Congenital Anomalies/Birth Defects Follow-Up of Patients after Adverse Events Investigator Follow-Up Sponsor Follow-Up Post-Study Adverse Events Expedited Reporting to Health Authorities, Investigators, Institutional Review Boards, | 89<br>89<br>90<br>90 |

| | 6.3 | Summaries of Treatment Group Comparability | 93 |
|-----|------------|-----------------------------------------------------|-----|
| | 6.4 | Efficacy Analyses | 93 |
| | 6.4.1 | Primary Efficacy Endpoint | 94 |
| | 6.4.2 | Secondary Efficacy Endpoints | 94 |
| | 6.5 | Safety Analyses | 96 |
| | 6.6 | Pharmacodynamic Analyses | 97 |
| | 6.7 | Pharmacokinetic Analyses | 97 |
| | 6.8 | Exploratory Analyses | 98 |
| | 6.9 | Interim Analyses | 98 |
| 7. | DATA COLL | ECTION AND MANAGEMENT | 98 |
| | 7.1 | Data Quality Assurance | 98 |
| | 7.2 | Electronic Case Report Forms | 99 |
| | 7.3 | Source Data Documentation | 99 |
| | 7.4 | Use of Computerized Systems | 99 |
| | 7.5 | Retention of Records | 100 |
| 8. | ETHICAL CO | ONSIDERATIONS | 100 |
| | 8.1 | Compliance with Laws and Regulations | 100 |
| | 8.2 | Informed Consent | 101 |
| | 8.3 | Institutional Review Board or Ethics Committee | 101 |
| | 8.4 | Confidentiality | 102 |
| | 8.5 | Financial Disclosure | 102 |
| 9. | | CUMENTATION, MONITORING, AND ATION | 102 |
| | 9.1 | Study Documentation | 102 |
| | 9.2 | Site Inspections | 103 |
| | 9.3 | Administrative Structure | 103 |
| | 9.4 | Publication of Data and Protection of Trade Secrets | 103 |
| | 9.5 | Protocol Amendments | 103 |
| 10. | REFERENC | ES | 105 |

# **LIST OF TABLES**

| Table 1 | Cycle 1 Mean (SD) Pharmacokinetic Parameters for Trastuzumab Emtansine Following Trastuzumab Emtansine Administration Every Three Weeks and Weekly in Study TDM3569g | 33 |
|---|---|---|
| Table 2 | Dose Reductions for Trastuzumab Emtansine (mBC Patients) | |
| Table 3 | Dose Reductions for Trastuzumab Emtansine (mGC Patients) | |
| Table 4 | Trastuzumab Emtansine Dose Modification: Total Serum Bilirubin | |
| Table 5 | Trastuzumab Emtansine Dose Modification: Serum ALT or AST | |
| Table 6<br>Table 7 | Adverse Event Severity Grading Scale | 83 |
| Table 8 | Adverse Event | 92 |
| | LIST OF FIGURES | |
| Figure 1 | Molecular Structure of Trastuzumab Emtansine | |
| Figure 2<br>Figure 3 | MMTV HER2 Fo5 Mammary Tumor Transplants Anti-tumor Activity of Trastuzumab Emtansine in | |
| Figure 4 | Combination with Capecitabine in NCI-N87 Overview of Study Design | 37 |
| Figure 5 | Overview of Study Design Overview of Phase I Dose Finding Study Design | 42<br>43 |
| Figure 6 | Algorithm for Continuation and Discontinuation of Trastuzumab Emtansine Based on Left Ventricular | |
| | Ejection Fraction Assessments in Patients | 76 |
| | LIST OF APPENDICES | |
| Appendix 1 | Schedule of Assessments | 109 |
| Appendix 2 | Pharmacokinetic Sampling for Phase I, Metastatic Breast and Gastric Cancer Patients | 119 |
| Appendix 3 | Response Evaluation Criteria in Solid Tumors (RECIST): Modified Excerpt from Original | 110 |
| | Publication | 120 |
| Appendix 4 | Instructions for Scans in the Event of Isotope | 120 |
| Appendix 5 | Shortage New York Heart Association Classification of | 132 |
| , appointed to | Functional Cardiac Capacity | 133 |

Date

# PROTOCOL ACCEPTANCE FORM

TITLE: PHASE I FOLLOWED BY PHASE II STUDY OF THE COMBINATION OF TRASTUZUMAB EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED OR METASTATIC GASTRIC CANCER PATIENTS


EUDRACT NUMBER: 2012-001547-46


MEDICAL MONITOR:

SPONSOR: F. Hoffmann-La Roche Ltd

I agree to conduct the study in accordance with the current protocol.

Principal Investigator's Name (print)

Please return a copy of the form to the contact provided below. Please retain the original for your study files.

Principal Investigator's Signature

#### **PROTOCOL SYNOPSIS**

TITLE: PHASE I FOLLOWED BY PHASE II STUDY OF THE COMBINATION OF

> TRASTUZUMAB EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED OR METASTATIC GASTRIC CANCER PATIENTS


2012-001547-46 **EUDRACT NUMBER:** 


PHASE:

INDICATION: HER2-positive metastatic breast and locally advanced or metastatic

gastric cancer

SPONSOR: F. Hoffmann-La Roche Ltd

#### **Objectives**

#### Phase I: Maximum Tolerated Dose Finding of Trastzumab Emtansine and Capecitabine in Metastatic Breast Cancer

#### Primary Objective

To determine the Maximum Tolerated Dose (MTD) of the combination of trastuzumab emtansine and capecitabine in metastatic breast cancer (mBC) patients

#### Secondary Objectives

- Pharmacokinetics (PK) of trastuzumab emtansine and metabolites and capecitabine
- · Safety of the combination of trastuzumab emtansine and capecitabine
- Overall Response Rate (ORR)

# Phase II: Exploration of Efficacy: mBC

#### **Primary Objective:**

ORR by investigator assessment

#### Secondary Objectives

- Safety profile of the combination at the dose established during Phase I
- Time to response (TTR)
- Duration of response (DoR)
- Time to progression (TTP)
- Time to treatment failure (TTF)
- Progression free survival (PFS)
- Clinical benefit rate (CBR)
- Overall survival (OS)

#### Phase I: MTD Finding of Trastzumab Emtansine and Capecitabine in Metastatic **Gastric Cancer**

#### Primary Objective

To determine the MTD of the combination of trastuzumab emtansine and capecitabine in metastatic gastric cancer (mGC) patients

- PK of trastuzumab emtansine and metabolites and capecitabine
- Safety of the combination of trastuzumab emtansine and capecitabine

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Overall Response Rate (ORR)

#### Study Design

#### **Description of Study**

This is an international, multicenter study.

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in HER2-positive mBC and locally advanced or mGC patients, using a Phase I design, followed by a Phase II single arm study to explore the efficacy of the combination in mBC patients. There will be no exploration of efficacy in the mGC cohort. Results from the Phase I in mGC will be used as supporting information for future studies in the indication (see Figure 4 in the protocol).

Cohort 1 (mBC) and Cohort 2 (mGC) will open sequentially during Phase I.

#### Phase I: MTD Finding, Cohort 1: mBC

Cohort 1 will open first with a 3 by 3 classical design. Cohort 1 will enroll patients with HER2-positive mBC. The dose tested of trastuzumab emtansine remains fixed at 3.6 mg/kg every 3 weeks and 3 dose levels of capecitabine administered twice daily on days 1 to 14 in cycles of 3 weeks will be tested. All patients will be treated until disease progression, intolerable toxicity, withdrawn consent, or death. All patients will be followed-up intolerable toxicity, withdrawn consent, death or up to a maximum of 2 years after the last patient was enrolled in the Phase II part of the study, whichever occurs first.

The rules for dose escalation are presented below.

If Dose level 1 is too toxic (dose limiting toxicity [DLT] >1/3 or >1/6) the combination may be considered unfeasible, recruitment will be closed and no other cohort will open. Patients who at that point experience response as per Response Evaluation Criteria for Solid Tumors (RECIST) will be offered the possibility to continue on trastuzumab emtansine as a single agent.

#### Dose Levels Explored in Phase I, Cohort 1:

Dose level 1: 750 mg/m<sup>2</sup> capecitabine twice daily (bid) + 3.6 mg/kg every three weeks (q3w) trastuzumab emtansine

Dose level 2: 850 mg/m<sup>2</sup> capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine

Dose level 3: 1000 mg/m² capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine

#### Phase II: Exploration of Efficacy, Cohort 1: mBC

Phase II will be conducted in mBC patients only.

Once the MTD in Cohort 1 is established, recruitment into this cohort will be extended to a total of 110 HER2-positive mBC patients for the Phase II part. Patients, who are on the MTD established in the Phase I part of the study, must re-consent to be enrolled into Phase II.

Patients will be treated until disease progression, intolerable toxicity withdrawn consent, or death. If capecitabine needs to be discontinued for any reason, trastuzumab emtansine may continue, and the patient will remain evaluable in the study. In case of discontinuation of trastuzumab emtansine, patients will be withdrawn from the study.

All patients will be followed up until disease progression, intolerable toxicity, withdrawn consent, death or up to a maximum of 2 years after the last patient was enrolled in the Phase II part of the study, whichever occurs first. Patients who have not progressed at that point in time may be enrolled into an extension study.

#### Phase I: MTD Finding, Cohort 2: mGC

Once the capecitabine MTD dose is established for Cohort 1, Cohort 2 will open, with a 3 by 3 classical design to enroll HER2-positive mGC patients. Trastuzumab emtansine will be administered weekly at the dose of 2.4 mg/kg and capecitabine will start at the MTD dose defined in Cohort 1, capecitabine dose level may be de-escalated.

All patients will be treated until disease progression, intolerable toxicity, withdrawn consent, or death. All patients will be followed-up until intolerable toxicity, withdrawn consent, death or up to a maximum of 2 years after the last patient was enrolled in the Phase II part of the study, whichever occurs first.

The dose levels for capecitabine will be the same as described in Cohort 1. Guidelines for dose escalation and de-escalation are as follows:

If MTD is defined at Dose Level 1 of 750 mg/m<sup>2</sup> bid:

Escalation will be to Dose Level 2 of 850 mg/m<sup>2</sup> bid.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

62

 De-escalation: if Dose Level 1 is not tolerated (>1/3 or >1/6 DLT), the combination will be considered not feasible.

If MTD defined at Dose Level 2 of 850 mg/m<sup>2</sup> bid:

- Escalation will be to Dose Level 3 of 1000 mg/m<sup>2</sup> bid
- De-escalation will be to Dose Level 1 of 750 mg/m<sup>2</sup> bid

If MTD defined at Dose Level 3 of 1000 mg/m<sup>2</sup> bid

- Escalation: There will be no escalation, MTD will be defined at Dose Level 3
- De-escalation will be to Dose Level 2 of 850 mg/m<sup>2</sup> bid

#### **Number of Patients**

Phase I: mBC

3 to 18 patients may be enrolled.

Phase II: mBC

Cohort 1 will be expanded to enroll 110 patients in total.

Phase I: mGC

3 to 18 patients may be enrolled.

#### **Target Population**

Phase I, Cohort 1: mBC

HER2-positive mBC patients will be enrolled.

Patients must have received at least one treatment regimen which includes a chemotherapy and trastuzumab agent.

Phase II, Cohort 1: mBC

HER2-positive mBC patients will be enrolled.

Patients must have received at least one treatment regimen which includes a chemotherapy and trastuzumab agent.

Phase I, Cohort 2: mGC

HER2-positive advanced mGC patients will be enrolled.

Patients must not have received prior chemotherapy for advanced/metastatic disease.

#### Inclusion Criteria:

#### For mBC Patients:

- 1. Age ≥ 18 years old
- 2. Signed informed consent prior to any study specific procedure
- 3. Able and willing to comply with protocol
- 4. Negative serum pregnancy test for women of childbearing potential (including pre menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential
- 5. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 6 months after the last dose of study treatment (see Section 5.2.4 in the protocol)
- 6. ECOG performance status of 0, 1, or 2
- 7. Blood:
- a) Platelet count > 100,000 cells/mm<sup>3</sup>
- b) International normalized ratio (INR) < 1.5 × the upper limit of normal (ULN)
- c) Absolute neutrophil count (ANC) > 1500 cells/mm<sup>3</sup>
- d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 8. Liver function:

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- a) Total bilirubin ≤ 1.5 × ULN except in patients with previously documented Gilbert's syndrome in which case total bilirubin ≤ 3 mg/dL is acceptable
- b) Serum glutamic oxaloacetic transaminase (SGOT)/AST and serum glutamic pyruvic transaminase (SGPT)/alanine transaminase (ALT)  $\leq$  2.5  $\times$  the ULN
- c) Alkaline phosphatase  $\leq$  2.5  $\times$  the ULN. Patients with hepatic and/or bone metastases: alkaline phosphatase  $\leq$  5  $\times$  the ULN
- 9. Renal function:
- a) Serum creatinine of < 177 µmol/L or calculated creatinine clearance (CL) > 50 mL/min. If urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24 hour urine collection and demonstrate ≤ 1 g of protein/24 hours
- 10 Cardiac function:
- a) Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (ECHO) or multiple gated acquisition (scan) (MUGA)
- 11. Histologically or cytologically confirmed breast cancer
- 12. HER2-positive disease immunohistochemistry (IHC) 3+ or *in situ* hybridization (ISH) positive
- Tumor block available or 15 slides for retrospective central confirmation of HER2positivity (central confirmation not necessary for enrolment)
- mBC with at least one measurable lesion according to RECIST
- 15. Disease progression on at least one regimen containing trastuzumab and chemotherapy
- 16. Patients must have recovered from previous treatments

#### For mGC Patients:

- Age ≥ 18 years old
- 2. Signed informed consent prior to any study specific procedure
- 3. Able and willing to comply with protocol
- 4. Negative serum pregnancy test for women of childbearing potential (including pre menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential
- 5. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 6 months after the last dose of study treatment (see Section 5.2.4 in the protocol)
- 6. ECOG performance status of 0, 1, or 2
- 7. Blood:
- a) Platelet count > 100,000 cells/mm<sup>3</sup>
- b) INR < 1.5 × the ULN
- c) ANC > 1500 cells/mm<sup>3</sup>
- d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 8. Liver function:
- a) Total bilirubin ≤ 1.5 × ULN except in patients with previously documented Gilbert's syndrome in which case total bilirubin ≤ 3 mg/dL is acceptable
- b) SGOT/AST and SGPT/ALT ≤ 2.5 × the ULN
- c) Alkaline phosphatase  $\leq$  2.5  $\times$  the ULN. Patients with hepatic and/or bone metastases: alkaline phosphatase  $\leq$  5  $\times$  the ULN
- 9. Renal function:

- a) Serum creatinine of < 177 µmol/L or calculated creatinine CL > 50 mL/min. If urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24 hour urine collection and demonstrate ≤ 1 g of protein/24 hours
- 10. Cardiac function:
- a) LVEF ≥ 50% by ECHO or MUGA
- 11. Histologically or cytologically confirmed GC
- 12. HER2-positive tumor (primary tumor or metastatic lesion), defined as either IHC 3+ alone or IHC 2+ in combination with ISH+, prospectively confirmed by a Sponsor-designated central laboratory prior to enrollment. ISH positivity is defined as a ratio of ≥ 2.0 for the number of HER2 gene copies to the number of signals for CEP17.
- a) Archival tumor samples obtained from primary or metastatic sites are acceptable.
- b) Invasive tumor for central confirmation of HER2 status is required.
- c) A formalin-fixed paraffin-embedded (FFPE) tissue block with at least 5 mm of invasive tumor for central confirmation is preferred.
  - If FFPE tissue blocks (or partial block) are unavailable due to country or site regulations, a minimum of 8 freshly cut unstained slides MUST be available for central review of HER2 status.
- 13. Inoperable locally advanced or mGC

#### **Exclusion Criteria:**

#### For mBC Patients:

- 1. Prior treatments before first study treatment:
- a) Investigational therapy within ≤ 28 days or 5 half lives, whatever is longest
- b) Hormonal therapy within 14 days
- c) Trastuzumab within 21 days
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received prior trastuzumab emtansine
- 3. Prior treatment with capecitabine
- 4. History of severe and unexpected reactions to fluoropyrimidine or with known hypersensitivity to fluorouracil
- 5. Related capecitabine contraindications:
- a) Treatment with sorivudine or its chemically related analogues, such as brivudine
- b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins
- 7. History of exposure to the following cumulative doses of anthracyclines:
- a) Doxorubicin or liposomal doxorubicin > 360 mg/m<sup>2</sup>
- b) Epirubicin > 900 mg/m<sup>2</sup>
- c) Mitoxantrone > 120 mg/m<sup>2</sup>
- d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 360 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 28 days of first study drug administration
- 9. Current peripheral neuropathy of Grade ≥ 3 per the NCI CTCAE, v4.0
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above
- 11. Current unstable ventricular arrhythmia requiring treatment
- 12. History of symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] Classes II–IV)

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
- 15. Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation
- 20. Current known active infection with HIV, hepatitis B, and/or hepatitis C virus
- a) For patients who are known carriers of hepatitis B virus (HBV), active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Lapatinib ≤ 14 days before first study drug administration
- 22. Previous radiotherapy for the treatment of unresectable, locally advanced/recurrent or mBC is not allowed if:
- The last fraction of radiotherapy has been administered within 14 days prior to first study drug administration
- b) More than 25% of marrow-bearing bone has been irradiated
- c) The patient has not recovered from any resulting acute toxicity to Grade ≤ 1 prior to first study drug administration

#### For mGC Patients:

- 1. Prior treatments before first study treatment:
- a) Investigational therapy within ≤ 28 days or 5 half lives, whatever is longest
- b) Hormonal therapy within 14 days
- c) Trastuzumab within 21 days
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received prior trastuzumab emtansine
- 3. Prior treatment with capecitabine
- 4. History of severe and unexpected reactions to fluoropyrimidine or with known hypersensitivity to fluorouracil
- 5. Related capecitabine contraindications:
- a) Treatment with sorivudine or its chemically related analogues, such as brivudine
- b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins
- 7. History of exposure to the following cumulative doses of anthracyclines:
- a) Doxorubicin or liposomal doxorubicin > 360 mg/m<sup>2</sup>
- b) Epirubicin > 900 mg/m<sup>2</sup>
- c) Mitoxantrone > 120 mg/m<sup>2</sup>
- d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 360 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 28 days of first study drug administration
- 9. Current peripheral neuropathy of Grade ≥ 3 per the NCI CTCAE, v4.0
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- 11. Current unstable ventricular arrhythmia requiring treatment
- 12. History of symptomatic CHF (NYHA Classes II-IV)
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
- 15. Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation
- 20. Current known active infection with HIV, hepatitis B, and/or hepatitis C virus
- a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Previous chemotherapy for advanced/metastatic disease
- a) Prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study

#### Length of Study

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to be 2 years for dose finding and the Phase II exploration of efficacy. All patients will be followed up until intolerable toxicity, withdrawn consent, death or up to a maximum of 2 years after the last patient was enrolled in the Phase II part of the study whichever occurs first. In case that Dose Level 1 is too toxic, the study may be terminated prematurely.

#### **End of Study**

Last Patient Last Visit (LPLV) as per definition is the last data collection point that can be either a clinic visit or a lab sample (see above length of study).

#### **Efficacy Outcome Measures**

Efficacy will be evaluated as per RECIST.

- Best overall response rate (BORR)
- Duration of response (DoR)
- Time to response (TTR)
- Time to progression (TTP)
- Time to treatment failure (TTF)
- Progression free survival (PFS)
- Clinical benefit rate (CBR)
- Overall survival (OS)

### **Safety Outcome Measures**

- Incidence and severity by NCI CTCAE version 4.0 of adverse events (AEs) and serious adverse events (SAEs)
- Cases and causes of death
- Laboratory parameters
- Left ventricular ejection fraction (LVEF)
- Treatment exposure

# Pharmacodynamic Outcome Measures

Hospital visit parameters.

#### **Pharmacokinetic Outcome Measures**

PK will be evaluated during Phase I for both trastuzumab emtansine and capecitabine (see Appendix 1, Schedule of Assessment in the protocol)

#### **Investigational Medicinal Products**

#### For mBC Patients:

Trastuzumab emtansine will be administered every 3 weeks at a dose of 3.6 mg/kg IV.

The total trastuzumab emtansine dose will be calculated based on the patient's weight on Day 1 of (or up to 3 days before) each cycle with no upper limit.

<u>Capecitabine</u> will be administered twice a day, orally for 14 days followed by a 7-day rest period at the dose levels 1–3 described in the 'Trial Design' section.

Capecitabine tablets should be swallowed with water within 30 minutes after a meal.

#### For mGC Patients:

<u>Trastuzumab emtansine</u> will be administered on Day 1 of a weekly cycle at the dose of 2.4 mg/kg IV.

The total trastuzumab emtansine dose will be calculated based on the patient's weight on Day 1 of (or up to 3 days before) each cycle with no upper limit.

<u>Capecitabine</u> will be administered twice a day, orally for 14 days followed by a 7-day rest period at the dose levels 1–3 described in the 'Trial Design' section.

Capecitabine tablets should be swallowed with water within 30 minutes after a meal.

#### **Non-Investigational Medicinal Products**

Not applicable.

#### **Statistical Analysis**

The study will include two phases and 2 cohorts:

Phase I, Cohort 1: mBC Dose Finding Cohort

Phase II, Cohort 1: mBC Exploration of Efficacy Cohort

Phase I, Cohort 2: mGC Dose Fining Cohort

During Phase I, the primary objective is reaching the MTD and establishing a safety profile.

There is no formal efficacy interim analysis.

Corresponding analyses as described in the protocol will be performed when all data for both cohorts and study phases are collected and cleaned

#### Analysis of primary and secondary endpoints:

#### **Analysis Populations:**

#### Phase I: MTD Finding: mBC Patients:

The main analysis population will be the safety population including all patients in this cohort who received at least one dose of study medication (trastuzumab emtansine and capecitabine) during this phase.

#### Phase II: Exploration of Efficacy: mBC Patients

The main analysis population for the efficacy analysis will be the intent-to-treat population (ITT) including all new patients enrolled in Phase II and patients from Cohort 1 who achieved the MTD level. The per-protocol (PP) population will include all ITT patients who have at least one post-baseline tumor assessment during the Phase II and no major protocol violations which will be defined in the statistical analysis plan. Safety parameters will be summarized for the safety population that includes all patients who received at least one dose of study medication in this part of the study.

#### Phase I: MTD Finding, mGC Patients:

The main analysis population will be the safety population including all patients in this cohort who received at least one dose of study medication (trastuzumab emtansine and capecitabine) during this phase.

#### Efficacy Endpoints:

#### Phase I: MTD Finding, mBC

The primary objectives are reaching the MTD and establishing a safety profile.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

ORR, as a main efficacy endpoint, will be assessed via BORR. The BOR is defined as the best response recorded from the date when the MTD is achieved until disease progression/recurrence (or death). The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### Phase II: Exploration of Efficacy: mBC

The primary efficacy endpoint for Phase II is the BOR as assessed by investigators. The BOR is defined as the best response recorded from the start of this Phase II until disease progression/recurrence (or death) or for patients who were involved in Phase I of the study: the best response from the date of the MTD reached until disease progression/recurrence or death. To be assigned a status of partial response (PR) or complete response (CR), i.e. to be a responder, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 28 days after the criteria for response are first met, i.e. patients need to have two consecutive assessments of PR or CR. This status will be assessed only for patients with measurable disease at baseline. Patients with non-measurable disease at baseline will be assessed for the time-to-event endpoints (e.g. PFS. OS. etc).

The number and proportions of responders and non-responders together with two-sided, 95% Clopper-Pearson confidence intervals will be presented. CBR will be summarized in a similar way.

#### The secondary endpoints for Phase II will be:

- Time to response (TTR)
- Duration of response (DoR)
- Time to progression (TTP)
- Time to treatment failure (TTF)
- Progression free survival (PFS)
- Clinical benefit rate (CBR)
- Overall survival (OS)

Estimates for the survivor function for the time-to-event variable such as TTR, DoR, TTP, TTF, PFS, and OS, will be obtained by using the Kaplan-Meier approach. CBR will be summarized in a similar way to the primary efficacy endpoint, BOR.

#### Phase I: MTD Finding: mGC

The primary objectives are reaching the MTD and establishing a safety profile.

Efficacy endpoints will be analysed in a similar way to Phase I: mBC.

#### **Safety Endpoints**

#### Phase I: MTD Finding: mBC

Safety parameters for this study part will be summarized by treatment dose. The summaries of AEs, SAEs, AEs that cause discontinuation from the study treatment will be analyzed in a similar way to AEs in Phase II. The summaries will include all patients who received at least one dose of study medication.

The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by MedDRA preferred term. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry, will be presented in shift tables of NCI-CTC grade at baseline versus worst grade during treatment for Phase I, Cohort 1, and overall.

LVEF will be summarized over time by means of mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

# Phase II: Exploration of Efficacy: mBC

# Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

69

Safety endpoints during Phase II will be assessed via: total AEs, AEs Grade ≥ 3, SAEs, premature withdrawal from study and study medication, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by MedDRA preferred term. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry, will be presented in shift tables of NCI-CTC grade at baseline versus worst grade during treatment for Phase II, Cohort 1 and overall.

LVEF will be summarized over time by means of mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### Phase I: MTD Finding: mGC

Safety parameters will be summarized in a similar way to Phase I: mBC.

#### Pharmacokinetic Analysis

The following pharmacokinetic parameters of trastuzumab emtansine and capecitabine (not limited to these listed) will be determined only in the Phase I part of the study in all patients who receive study treatment using either non-compartmental and/or population methods, if data allow:

- Serum concentrations of trastuzumab emtansine (conjugate) and total trastuzumab
- Plasma concentrations of DM1, capecitabine and its active metabolite 5-fluorouracil (5-FU)
- Total exposure (AUC)
- C<sub>max</sub>
- · Clearance (CL)
- Volume of distribution (V<sub>d</sub>)
- Terminal half-life (T<sub>1/2</sub>)

All PK parameters will be listed and tabulated by treatment dose and by Cohort. Descriptive summary statistics including arithmetic mean, geometric mean (e.g. AUC and  $C_{\text{max}}$ ), median, range, standard deviation (SD) and coefficient of variation will be presented for each Cohort. Nonlinear mixed effects modeling will be also used but details will be presented in the statistical anal analysis plan.

### **Exploratory Analyses**

Subgroup analysis for BOR, safety (AEs, SAEs and AE with Grade ≥ 3) in Phase II will be presented for: elderly *versus* younger patients, patients with ECOG 0–1 *versus* ECOG 2. More details will be presented in the statistical analysis plan.

#### Pharmaceconomic Endpoint

The number of hospital visits, number of days admitted, and type of visits (emergency department versus inpatient care) will be collected and compared. The reason for admission (disease progression *versus* AE) will also be assessed.

# **Determination of Sample Size**

#### Sample Size for Phase I: MTD Finding: mBC

This part will be based on a classical 3 by 3 Phase I design. From 3 to 18 patients might be enrolled in Cohort 1. There is no formal sample size estimation for this part.

# Sample Size for Phase II: Exploration of Efficacy: mBC

Assuming a preferable BORR of 75% to 80% in Cohort 1 (mBC patients) and aiming for a precision of 8-10%, lower limit of 95% confidence interval of at least 65%, a total of 100 patients would need to be evaluable for Cohort 1.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Table 1: Sample Size Estimation

| Total number of patients is 100 (Phase II) | |
|---|---|
| Number of Patients/ Response | 95% Clopper-Pearson<br>Confidence Intervals |
| 75 patients (75%) | 65% - 83 % |
| 80 patients (80%) | 71% - 87% |
| Total number of patients adjusted for 10% withdrawal rate is 110 patients | |

For example, the observed BOR of 75% could be estimated to be within 65% and 83% with a probability of 95% (Clopper-Pearson exact confidence intervals). Adjusting for a withdrawal rate of approximately 10%, 110 patients will be enrolled in this phase.

The BOR rate of 75% is chosen based on the previously published data with trastuzumab and capecitabine (see protocol for reference)

The estimation of Sample Size is performed by Nquery and SAS programs.

#### Sample Size for Phase I: MTD Finding: mGC

This part will be based on a classical 3 by 3 Phase I design. From 3 to 18 patients might be enrolled in Cohort 2. There is no formal sample size estimation for this part.

# **LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS**

| Abbreviation | Definition |
|------------------|------------------------------------------------|
| ADL | activities of daily living |
| AE | adverse event |
| ADC | antibody-drug conjugate |
| ALT | alanine transaminase |
| ANC | absolute neutrophil count |
| aPTT | activated partial thromboplastin time |
| ARDS | acute respiratory distress syndrome |
| AST | aspartate transaminase |
| AUC | area under the serum concentration-time curve |
| BC | breast cancer |
| bid | twice daily |
| BML | below measurable limit |
| BOR | best overall response |
| BORR | best overall response rate |
| BUN | blood urea nitrogen |
| CBR | clinical benefit rate |
| CHF | congestive heart failure |
| CI | confidence interval |
| CL | clearance |
| C <sub>max</sub> | maximum concentration |
| CR | complete response |
| CRO | contract research organization |
| CSR | clinical study report |
| СТ | computed tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DLT | dose limiting toxicity |
| DoR | duration of response |
| DPD | dihydropyrimidine dehydrogenase |
| 5`DFUR | 5'-deoxy-5-fluorouridine |
| 5`FU | 5-fluoruracil |
| EC | Ethics Committee |
| ECG | electrocardiogram |
| ECHO | echocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| EEA | European economic area |
| EU | European Union |

| FDA | Food and Drug Administration |
|--------|---------------------------------------------------------------|
| FISH | fluorescence in situ hybridization |
| GC | gastric cancer |
| GCP | Good Clinical Practice |
| GEJ | gastroesophageal junction |
| HER2 | human epidermal growth factor receptor 2 |
| HIPAA | Health Insurance Portability and Accountability Act |
| HR | hazard ratio |
| HIV | human influenza virus |
| ICH | International Conference on Harmonisation |
| IHC | immunohistochemistry |
| IMP | investigational medicinal product |
| IND | Investigational New Drug (application) |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| ITT | intent-to-treat |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| IxRS | interactive voice/web recognition system |
| LVEF | left ventricular ejection fraction |
| mBC | metastatic breast cancer |
| mGC | metastatic gastric cancer |
| MRI | magnetic resonance imaging |
| MTD | maximum tolerated dose |
| MUGA | multiple-gated acquisition (scan) |
| NCI | National Cancer Institute |
| NE | not evaluable |
| ORR | overall response rate |
| os | overall survival |
| PD | pharmacodynamic/progressive disease |
| PET | positron emission tomography |
| PFS | progression free survival |
| PK | pharmacokinetic |
| PP | per-protocol |
| PR | partial response |
| QTcF | heart rate-corrected QT interval using the Fridericia formula |
| q3w | every 3 weeks |
| qw | weekly |
| RECIST | Response Evaluation Criteria for Solid Tumors |
| L | |

| SAE | serious adverse event |
|------------------|-----------------------------------------|
| SGOT | serum glutamic oxaloacetic transaminase |
| SD | standard deviation |
| SGPT | serum glutamic pyruvic transaminase |
| SWFI | sterile water for injection |
| T <sub>1/2</sub> | terminal half-life |
| TTF | time to treatment failure |
| TTP | time to progression |
| TTR | time to response |
| ULN | upper limit of normal |
| V | volume of distribution |
| WBC | white blood cells |
| WHO | World Health Organization |

# 1. BACKGROUND

# 1.1 BACKGROUND ON DISEASE

# 1.1.1 HER2-Positive Breast Cancer, Metastatic Breast Cancer

Breast cancer (BC) is the most common cancer in women worldwide, both in the developed and the developing world (WHO, World Health Statistics. 2011), with approximately 1.38 million new cases diagnosed in 2008. It is also the leading cause of cancer death in females, accounting for 458,400 deaths (14% of all cancer deaths) in 2008 (Jemal et al. 2011). Almost 100,000 of these BC-related deaths occurred in patients whose tumors overexpressed human epidermal growth factor receptor 2 (HER2) receptors. Metastatic breast cancer (mBC) is incurable, with the primary goal of treatment to extend life and palliate symptoms while preserving quality of life.

The HER tyrosine kinase receptor family is comprised of four receptors: HER1, HER2, HER3, and HER4. These receptors are important mediators of cell growth, survival, and differentiation (Sundaresan et al. 1999). Activation of HER receptors leads to receptor dimerization and cell signaling through the PI3-kinase/AKT pathway for promotion of tumor cell survival and through the mitogen-activated protein kinase pathway for cellular proliferation.

Overexpression of HER2 is observed in approximately 15–20% of human BCs. Several lines of scientific and clinical evidence support a direct role for HER2 overexpression in the aggressive growth and poor clinical outcomes associated with these tumors (Slamon et al. 1987). The development of trastuzumab in the 1990s provided women with HER2-overexpressing tumors with a markedly better outcome than was possible with chemotherapy alone. Increases in response rate, response duration, and progression free survival (PFS) were associated with a 5-month survival advantage when trastuzumab was given in the first-line metastatic setting, as demonstrated in the initial Phase III trial (Slamon et al. 2001).

For patients with HER2-positive mBC, the combination of trastuzumab and a taxane is a globally accepted first-line treatment, based on the survival advantage demonstrated in two large pivotal trials (Slamon et al. 2001; Marty et al. 2005). However, virtually all patients with HER2-positive mBC develop progressive disease (PD) and require additional therapies. Importantly, such tumors continue to express high levels of HER2 (Spector et al. 2005), and neither the process of internalization nor the level of surface expression is altered when HER2 is bound by trastuzumab (Austin et al. 2004). HER2-directed combination therapy beyond progression for HER2-positive mBC is an accepted palliative treatment approach.

An accepted example of second-line therapy for HER2-positive mBC therapy is lapatinib in combination with capecitabine as a treatment for patients who have received trastuzumab and a taxane for advanced disease. In a Phase III trial involving patients with advanced HER2-positive BC previously treated with an anthracycline, a taxane, and trastuzumab, the addition of lapatinib to

capecitabine resulted in an increased response rate (24% *versus* 14%) and time to disease progression (6.2 months *versus* 4.3 months) (Geyer et al. 2006).

Capecitabine (Xeloda®) in combination with docetaxel for treatment of patients with locally advanced or mBC after failure of cytotoxic chemotherapy, including an anthracycline was studied in a multicenter, randomized, controlled Phase III clinical trial (SO14999). In this trial, 255 patients were randomized to treatment with capecitabine (1250 mg/m² twice daily (bid) for 2 weeks followed by a 1-week rest period) and docetaxel (75 mg/m<sup>2</sup> as a 1-hour intravenous [IV] infusion every 3 weeks). A total of 256 patients were randomized to treatment with docetaxel alone (100 mg/m<sup>2</sup> as a 1-hour IV infusion every 3 weeks). Survival was superior in the capecibabine plus docetaxel combination arm (p = 0.0126). Median survival was 442 days (capecitabine plus docetaxel) versus 352 days (docetaxel alone). The overall objective response rates in the all-randomized population (investigator assessment) were 41.6% (capecitabine plus docetaxel) versus 29.7% (docetaxel alone); p = 0.0058. Time to progression (TTP) of disease or number of deaths was superior in the capecitabine plus docetaxel combination arm (p < 0.0001). The median TTP was 186 days (capecitabine plus docetaxel) versus 128 days (docetaxel alone).

Two multicenter Phase II clinical trials were conducted to determine the use of capecitabine monotherapy for treatment of patients with locally advanced or mBC after failure of a taxane and an anthracycline-containing chemotherapy regimen or for whom further anthracycline therapy is not indicated. In these trials, a total of 236 patients were treated with capecitabine (1250 mg/m² bid for 2 weeks followed by 1-week rest period). The overall objective response rates (investigator assessment) were 20% (first trial) and 25% (second trial). The median TTP was 93 and 98 days. Median survival was 384 and 373 days (Blum et al. 1999; Blum et al. 2001).

# 1.1.2 HER2-Positive Locally Advanced or Metastatic Gastric Cancer

Gastric cancer (GC) remains one of the most common malignancies in the world with an estimated 989,600 new cases in 2008 (Jemal et al. 2011). GC also continues to be a deadly disease; it is the second leading cause of cancer-related death accounting for 738,000 deaths (9.7% of all cancer deaths) worldwide in 2008 (Ferlay et al. 2010). The only potentially curative treatment for GC is complete resection of localized disease. The overall 5-year survival for all cases, regardless of initial stage at diagnosis, is less than 25% (Catalano et al. 2005; Faivre et al. 1998; Parkin et al. 2005; Power et al. 2010). Among patients with localized disease who undergo curative surgery, approximately 40–60% will have disease recurrence. Patients with unresectable disease due to locally advanced growth or metastatic spread have the poorest prognosis, with an overall 5-year survival in the range of 3–15% (De Vivo et al. 2000; Ries et al. 2008; Power et al. 2010).

Whereas HER2 overexpression is associated with a poor prognosis in BC, the prognostic significance of HER2 overexpression in GC is not fully defined.

Studies of HER2 positivity rates in GC have shown a broad variation of HER2 positivity ranging from 6.8–34.0% for immunohistochemistry (IHC) and 7.1–42.6% for fluorescence *in situ* hybridization (FISH) techniques (Hofmann et al. 2008; Tanner et al. 2005). In a recent study, HER2 positivity was shown in 17% of resected esophageal adenocarcinomas and was significantly associated with lower tumor grade, less invasiveness, fewer malignant nodes, and the presence of adjacent Barrett's esophagus (Yoon et al. 2012).

In the ToGA trial (study BO18255), a global, Phase III study of trastuzumab plus chemotherapy as first-line treatment for advanced HER2-positive GC, an overall HER2-positivity rate of 22.1% was observed (810/3667 evaluable samples), which is comparable to BC. A higher HER2-positivity rate was seen in adenocarcinoma of the gastroesophageal junction (GEJ) than in the stomach (33.2% *versus* 20.9%), and intestinal type GCs showed a significantly higher HER2-positivity rate than diffuse or mixed-type tumors (intestinal: 32.2%, diffuse: 6.1%, mixed: 20.4%) (Albarello et al. 2011; Bang et al. 2010).

In the ToGA trial (study BO18255), the addition of trastuzumab to chemotherapy (capecitabine or fluorouracil combined with cisplatin) for the treatment of patients with HER2-positive (defined as IHC 3+ or FISH positive), inoperable, locally advanced or recurrent and/or metastatic adenocarcinoma of the stomach or GEJ resulted in an increase in the median overall survival ([OS]; 13.8 months *versus* 11.1 months, hazard ratio [HR] 0.74, p = 0.0046), objective response rate (47% *versus* 35%), PFS (6.7 *versus* 5.5 months), and TTP (7.1 *versus* 5.6 months) compared with chemotherapy alone (Bang et al. 2010).

# 1.2 BACKGROUND ON STUDY DRUGS

### 1.2.1 TRASTUZUMAB EMTANSINE

Trastuzumab emtansine (also known as T-DM1, see Figure 1) is a novel antibody-drug conjugate (ADC) that is specifically designed for the treatment of HER2-positive malignancies. Trastuzumab emtansine is composed of trastuzumab, a humanized monoclonal antibody directed against the extracellular region of HER2; an average of 3.5 molecules of DM1 (maytansinoid), an anti-microtubule agent derived from maytansine; and the thioether linker maleimidylmethyl cylcohexane-1-carboxylate, which is used to conjugate each molecule of DM1 to trastuzumab. DM1 is a highly potent drug synthesized from maytansinol that binds β tubulin to inhibit tubulin polymerization. It binds to tubulin competitively with vinca alkaloids, but is 20-100 times more potent than vincristine in its cytotoxic effect against tumor cell lines. Its parent molecule, maytansine, has been studied in approximately 800 cancer patients in the 1970s and 1980s, with responses seen in patients with breast and lung cancer (Junttila et al. 2011; Issell, Crooke 1978). However, because of its narrow therapeutic index and the observed gastrointestinal toxicity of the free drug, it was not developed further as a therapeutic option (Cassady et al. 2004; Cabanillas et al. 1979).

Figure 1 Molecular Structure of Trastuzumab Emtansine



DM1 = Derivative of Maytansine, a microtubule destabilizing agent MW = Molecular weight

Similar to trastuzumab, trastuzumab emtansine recognizes an epitope in the extracellular domain of HER2 and binds to HER2 with a similar affinity. Following antigen specific binding of trastuzumab emtansine to HER2, the complex of receptor and ADC is internalized, whereupon DM1-containing catabolites are released into the cytosol following proteolytic cleavage of the antibody in lysosomes (Erickson et al. 2006). Binding of these DM1-containing species to β-tubulin inhibits tubulin polymerization resulting in cell death (Cassady et al. 2004).

In addition to targeting delivery of DM1 to HER2-overexpressing tumor cells, trastuzumab emtansine retains the anti-tumor activities of trastuzumab, including suppression of HER2 signaling pathways that confer a proliferative and survival advantage to cells, and the flagging of cells for destruction through antibody-dependent cell cytotoxicity (Junttila et al. 2011).

Completed and ongoing Phase I and II single arm studies of trastuzumab emtansine have shown clinical activity. Furthermore, low levels of DM1 in systemic circulation supported the stability of the linker (Shen et al. ASCPT 2011). The randomized Phase II study TDM4450g described in Section 1.2.1.4 showed a significant improvement in PFS with a HR 0.59 p=0.0353 and a favorable safety profile. A Phase III study (TDM4370g) is underway comparing trastuzumab emtansine to HER2-targeted combination therapy (capecitabine and lapatinib) for patients with mBC who had received prior trastuzumab and taxane therapies.

Data from clinical trials of trastuzumab emtansine that are relevant to the design of the current trial are summarized below. Please refer to the

trastuzumab emtansine Investigator's Brochure for further information on all of the completed and ongoing trastuzumab emtansine studies.

# 1.2.1.1 Study TDM3569g

Study TDM3569g was a Phase I, dose-escalation study that evaluated the safety and efficacy of trastuzumab emtansine as a single agent in 52 patients with HER2-positive mBC, whose disease progressed on a trastuzumab-containing chemotherapy regimen. The study was completed on 11 June 2009, with a total of 52 patients treated; 24 patients received trastuzumab emtansine every 3 weeks (q3w); 28 patients received trastuzumab emtansine on a weekly (qw) schedule.

On the q3w dosing schedule, dose limiting toxicities of Grade 4 thrombocytopenia, were seen in 2 of 3 patients treated at 4.8 mg/kg. Therefore, 3.6 mg/kg was determined to be the maximum tolerated dose (MTD) of trastuzumab emtansine given q3w, and the cohort was expanded to 15 patients. On the basis of these data, the recommended dose schedule for the Phase II studies was 3.6 mg/kg q3w. On the qw schedule, 2.4 mg/kg was identified as the MTD (Krop et al. 2008).

Treatment with trastuzumab emtansine was well tolerated, and toxicity was generally mild, reversible, and non-cumulative. No drug-related cardiac toxicity was noted.

Trastuzumab emtansine administration demonstrated considerable activity in this Phase I study. The confirmed overall response rate (ORR) in patients with measurable disease at the 3.6 mg/kg q3w schedule was 44% (4 of 9 patients), as assessed by investigators. The median PFS among the 15 patients receiving 3.6 mg/kg q3w was 10.4 months.

#### 1.2.1.2 Study TDM4258g

Study TDM4258g was a Phase II study that evaluated the safety and efficacy of trastuzumab emtansine administered at a dose of 3.6 mg/kg (IV) q3w in HER2-positive mBC patients who had progressed on previous HER2-directed therapy and conventional chemotherapy.

The primary objectives for this study were: 1) to assess the ORR (by independent radiologic review) associated with trastuzumab emtansine 3.6 mg/kg IV q3w, and 2) to characterize the safety and tolerability of trastuzumab emtansine at this dose.

The study was activated on 20 July 2007, and enrollment was completed (n = 112) on 31 July 2008. The final analysis of ORR was performed with a data cut-off date of 25 June 2009, 11 months after the last patient was enrolled. The reported ORR in all patients was 37.5% (95% confidence interval [CI], 28.6%, 46.6%) by investigator assessment and 25.9% (95% CI, 18.4%, 34.4%) by Independent Review Committee (IRC). The clinical benefit rate ([CBR]; defined as complete response [CR], partial response [PR], or stable disease for >6 months) was 46.3% by investigator assessment and 39.3% by independent review. The median PFS was 4.6 months as assessed by both the investigators and the IRC. In the subset of patients whose archival

primary tumors were retrospectively confirmed to be HER2-positive (74 of 95 patients with submitted tumor samples), the ORR was 33.8% by independent review and 47.3% based on investigator assessment.

The most common adverse events (AEs) (occurring in  $\geq$ 20% of patients) were fatigue (65.2%), nausea (50.9%), headache (40.2%), epistaxis (35.7%), pyrexia (34.8%), constipation (30.4%), cough (27.7%), hypokalemia (26.8%), diarrhea (25.9%), vomiting (24.1%), arthralgia (22.3%), pain in extremity (22.3%), anemia (20.5%), and dyspnoea (20.5%). Most of these AEs were Grade 1–2. The three most common Grade 3–4 AEs observed in this trial were hypokalemia (8.9%), thrombocytopenia (8.0%), and fatigue (4.5%). There was one reported Grade 5 event in a patient who died of respiratory failure attributed by the investigator to underlying disease. No Grade  $\geq$ 3 left ventricular systolic dysfunction events (symptomatic congestive heart failure [CHF] and/or left ventricular ejection fraction [LVEF] of <40%) were observed.

# 1.2.1.3 Study TDM4374g

Study TDM4374g was a Phase II, single arm study of trastuzumab emtansine administered at 3.6 mg/kg by IV infusion q3w to patients with HER2-positive mBC. Patients must have received an anthracycline, trastuzumab, a taxane, lapatinib, and capecitabine given in the neoadjuvant, adjuvant, or metastatic setting or as treatment for locally advanced disease. Patients must have been treated with two HER2-directed therapies in the metastatic or locally advanced setting and have progressed on their most recent treatment.

The primary objectives of this study were: 1) to assess the ORR as assessed by an independent review using the modified Response Evaluation Criteria for Solid Tumors (RECIST) v. 1.0, and 2) to characterize the safety and tolerability of this trastuzumab emtansine regimen in the aforementioned patient population. The study was activated on 2 May 2008, and enrollment was complete on 2 April 2009. A total of 110 patients were enrolled and treated in the study.

An efficacy analysis (data cut-off date: 21 June 2010) with a median follow-up of 17.4 months demonstrated an ORR (complete and PR) of 34.5% (95% CI: 26.1–43.9%; 38 of 110 patients) by independent review and 32.7% (95% CI: 24.1–42.1%; 36 patients) by investigator assessment. The CBR was 48.2% by independent review and 46.4% by investigator assessment. The median duration of response (DoR) and PFS by independent review was 7.2 months and 6.9 months, respectively. In the subset of patients whose archival primary tumors were retrospectively confirmed to be HER2-positive (80 of 95 patients with submitted tumor samples), the ORR was 41.3% by independent review and 40.0% based on investigator assessment.

The most common AEs (occurring in ≥20% of patients) were fatigue (61.8%), thrombocytopenia (38.2%), nausea (37.3%), increased aspartate transaminase (AST, 26.4%), constipation (23.6%), pyrexia (22.7%), epistaxis (22.7%), headache (21.8%), hypokalemia (20.9%), decreased appetite (20.9%), dry mouth (20.0%), and anemia (20.0%). Most of these AEs were Grade 1–2. Fifty-two patients (47.3%) experienced at least one Grade ≥3 AE, the most common being thrombocytopenia (9.1%) and fatigue (4.5%). Serious

AEs were recorded by 28 patients (25.5%), the most common being cellulitis (3.6%), pyrexia (2.7%), and pneumonia (2.7%). One patient recorded a Grade 5 AE of hepatic dysfunction, which was recorded as possibly related to trastuzumab emtansine. The patient had pre-existing non-alcoholic fatty liver disease as well as multiple other co-morbidities, including renal insufficiency.

### 1.2.1.4 Study TDM4450g

This was a randomized, multicenter, Phase II study of the efficacy and safety of trastuzumab emtansine *versus* trastuzumab plus docetaxel in patients with metastatic HER2-positive breast cancer who had not received prior chemotherapy for metastatic disease. This study completed enrollment in December 2009 (n = 137). The primary objectives were to assess the efficacy of trastuzumab emtansine compared with the combination of trastuzumab and docetaxel, as measured by PFS based on investigator tumor assessments, and to characterize the safety of trastuzumab emtansine compared with the combination of trastuzumab and docetaxel in this population. Secondary endpoints included ORR, survival, and DoR.

The data cut-off date was 15 November 2010. Seventy patients were randomized to the control arm and 67 patients to the trastuzumab emtansine arm. The median duration of follow-up was 13.5 months for the control arm and 13.8 months for the trastuzumab emtansine arm.

As of 15 November 2010, the PFS was 14.2 months in the trastuzumab emtansine arm versus 9.2 months in the trastuzumab plus docetaxel arm. The HR for PFS was 0.594 (95% CI: 0.364-0.968; p = 0.0353). The ORR in the trastuzumab emtansine arm was 64.2% (95% CI: 51.8-74.8%) compared with 58.0% (95% CI: 45.5-69.2%) in the control arm (based on 69 evaluable patients). The CBR was 74.6% (95% CI: 63.2-84.2%) in the trastuzumab emtansine arm versus 81.2% (95% CI: 70.7–89.1%) in the trastuzumab plus docetaxel arm (based on 69 evaluable patients). Based on safety data analyzed at the data cut-off date, single agent trastuzumab emtansine appears to have a favorable overall safety profile compared with trastuzumab and docetaxel in first-line mBC. The incidence of Grade ≥3 AEs in the control arm (89.4%; n = 66) was nearly twice that of trastuzumab emtansine (46.4%; n = 69). The rates of serious AEs for both arms were similar (control arm 25.8% versus trastuzumab emtansine 18.8%). One patient in the trastuzumab emtansine group died as a result of an AE (sudden death). This patient was randomized to receive trastuzumab plus docetaxel but mistakenly received a single dose of 6 mg/kg trastuzumab emtansine instead of 6 mg/kg trastuzumab. One patient in the trastuzumab plus docetaxel group died due to cardiopulmonary failure. With respect to cardiotoxicity, based on local assessments of LVEF, trastuzumab emtansine was not associated with an increase in cardiotoxicity compared with trastuzumab plus docetaxel.

# 1.2.1.5 Study TDM4688g

The effect of trastuzumab emtansine (3.6 mg/kg q3w) on the QT interval in patients with HER2-positive recurrent locally advanced breast cancer or mBC was evaluated in study TDM4688g, and had no meaningful effect on the corrected QT interval in these patients. At Cycle 1 Day 1, 15 minutes post-

**Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 1

infusion, the baseline-adjusted average heart rate-corrected QT interval using the Fridericia formula (QTcF) increased by 1.2 ms on average. By 60 minutes post-infusion, the baseline-adjusted average QTcF interval decreased by 1.0 ms on average, and by Day 8 of Cycle 1, the baseline-adjusted average QTcF interval decreased by 4.0 ms on average. By Cycle 3 Day 1, prior to trastuzumab emtansine infusion, the average QTcF interval had reverted back to baseline on average. Following the third infusion of trastuzumab emtansine, the baseline-adjusted average QTcF interval at both the 15 minute and the 60 minute post-infusion time points was increased by an average of 4.7 ms. No patient exhibited an average change in QTcF interval from baseline exceeding 30 ms at any of the protocol-specified time points.

The relationship between trastuzumab emtansine pharmacokinetic (PK) and electrocardiogram (ECG) data was also assessed. While there appears to be a trend between trastuzumab emtansine drug concentration and its effect on QT interval, at the observed concentration ranges of trastuzumab emtansine, DM1, and total trastuzumab, there is reasonable assurance that the true increase in mean baseline-adjusted average QTcF does not exceed 5 ms. Moreover, because trastuzumab emtansine, total trastuzumab, and DM1 achieve steady state levels by Cycle 3, the likelihood of progressively longer QTcF with repeated trastuzumab emtansine dosing is low.

In this study, an ORR of 25.5% (95% CI: 15.2–38.5%) was assessed by the investigator; no independent review was performed in this study. The CBR was 39.2% (95% CI: 25.8–53.1%), and the median PFS was 4.3 months (95% CI: 4.0–6.7).

# 1.2.1.6 Phase III Study TDM4370g

Roche is conducting a randomized, open-label Phase III trial (TDM4370g) of single agent trastuzumab emtansine *versus* lapatinib and capecitabine in HER2-positive locally advanced unresectable BC or mBC patients who have received a prior taxane and trastuzumab therapy and have documented disease progression. The study is ongoing, enrollment is completed, and 991 patients have been enrolled.

Patients are randomized in a 1:1 ratio to trastuzumab emtansine or capecitabine plus lapatinib.

Trastuzumab emtansine is administered at 3.6 mg/kg IV every three weeks. The control arm treatment is capecitabine at 1000 mg/m² as oral doses bid on Days 1–14 of a q3w cycle plus oral lapatinib 1250 mg/day given as continuous dosing. Study treatment is discontinued based on disease progression (as assessed by the investigator), unmanageable toxicity or study termination by Roche/Genentech.

PFS and OS are investigated as co-primary endpoints in this study with PFS based on modified RECIST (Therasse et al. 2000) and conducted by the IRC. An additional tumor assessment of PFS is performed after investigator-documented disease progression. Furthermore ORR, DoR, and CBR are included, on the basis of both investigator and independent review of tumor assessments, as key secondary endpoints.

This trial has met its co-primary endpoint of improving PFS (by independent review committee) compared to those who received the combination of lapatinib and capecitabine.

PFS was 9.6 months in the trastuzumab emtansine arm versus 6.4 months in the lapatinib and capecitabine arm. OS has not yet been reached in the trastuzumab emtansine arm while in the control arm the OS was 23.3 months. The HR for PFS was 0.650 (95% CI: 0.55, 0.77; p = 0.0001). The ORR in the trastuzumab emtansine arm was 43.6% (95% CI: 38.6, 48.6) compared with 30.8% (95% CI: 26.3, 35.7) in the control arm (based on 786 evaluable patients). Based on safety data analyzed at the data cutoff date, single-agent trastuzumab emtansine appears to have a favorable overall safety profile compared with lapatinib and capecitabine in mBC. The incidence of Grade  $\geq$ 3 AEs in the control arm (56.9%; n = 488) was 278; that of trastuzumab emtansine (40.8%; n = 490) was 200. The rates of SAEs for both arms were similar (control arm 18% versus trastuzumab emtansine 15.5%).

It is concluded that overall, there is no concern regarding the clinical safety of trastuzumab emtansine based on the currently available data.

#### 1.2.1.7 Pharmacokinetics

The PK of trastuzumab emtansine and its analytes (total trastuzumab and DM1) were characterized in one Phase I study (TDM3569g) and three Phase II studies (TDM4258g, TDM4374g, and TDM4688g).

For study TDM3569g, the final PK parameter estimates based on non-compartmental PK analysis for q3w and qw regimens of trastuzumab emtansine administration are presented in Table 1.

Table 1 Cycle 1 Mean (SD) Pharmacokinetic Parameters for Trastuzumab Emtansine Following Trastuzumab Emtansine Administration Every Three Weeks and Weekly in Study TDM3569g

| Dose | No. of | C <sub>max</sub> | AUC <sub>inf</sub> | T <sub>1/2</sub> | V | CL |
|---|---|---|---|---|---|---|
| (mg/kg) | Patients | (µg/mL) | (day µg/mL) | (day) | (mL/kg) | (mL/day/kg) |
| Every 3 Week Dosing | | | | | | |
| 0.3 | 3 | 9.6 (1.7) | 14.5 (3.4) | 1.3 (0.2) | 35.7 (7.5) | 21.1 (4.5) |
| 0.6 | 1 | 13.3 | 24.5 | 1.3 | 43.8 | 24.5 |
| 1.2 | 1 | 20.3 | 42.9 | 1.3 | 51.8 | 27.8 |
| 2.4 | 1 | 76.3 | 330.0 | 2.2 | 30.7 | 7.2 |
| 3.6 | 15 | 76.2 (19.1) | 300.3 (65.8) | 3.1 (0.7) | 58.4 (12.4) | 12.7 (3.6) |
| 4.8 | 3 | 130.3 (7.8) | 673.0 (12.2) | 4.1 (0.7) | 41.2 (6.2) | 7.1 (0.1) |
| Weekly Dosing | | | | | | |
| 1.2 | 3 | 29.6 (5.7) | 76.2 (10.4) | 2.3 (0.6) | 47.5 (6.0) | 15.9 (2.4) |
| 1.6 | 3 | 34.3 (4.8) | 130.3 (39.7) | 3.4 (0.8) | 59.8 (16.6) | 13.0 (3.4) |
| 2.0 | 3 | 48.0 (9.6) | 175.0 (41.0) | 3.1 (0.3) | 51.0 (8.1) | 11.8 (2.4) |
| 2.4 | 16 | 54.8 (12.6) | 198.5 (54.5) | 3.3 (1.1) | 55.4 (13.0) | 13.1 (4.1) |
| 2.9 | 3 | 78.1 (33.9) | 212.0 (39.0) | 2.9 (0.5) | 57.7 (2.2) | 14.0 (2.6) |

AUC<sub>inf</sub> = area under the serum concentration-time curve from time 0 extrapolated to infinity;  $C_{max}$  = maximum serum concentration; CL = clearance; SD = standard deviation;  $T_{1/2}$  = terminal half-life; V = volume of distribution.

Dose intensity, defined as percentage of the planned trastuzumab emtansine dose that was actually received, was higher with the 3.6 mg/kg q3w regimen (median 99.7%, range 88%–106%) than with the 2.4 mg/kg qw schedule (median 82%, range 54%–101%). However, since the PK of trastuzumab emtansine is linear at doses ≥2.4 mg/kg, an almost 2-fold higher cumulative dose can be administered within a q3w cycle with a 2.4 mg/kg qw regimen compared to 3.6 mg/kg q3w (Krop et al. 2009, Krop et al 2010).

Based on a population PK analysis, trastuzumab emtansine has a consistent PK profile with low inter-individual variability (21–48%) in PK parameters among patients with mBC. Greater baseline tumor burden and lower serum albumin levels, potential indicators of disease severity, resulted in small increases (<13%) in trastuzumab emtansine clearance (CL). However, trastuzumab emtansine PK was not affected by baseline residual trastuzumab (from prior treatment) or by differences in serum concentrations of HER2 extracellular domain (Gupta et al. 2011).

An aggregate PK assessment of trastuzumab emtansine was done with samples from studies TDM3569g, TDM4258g, TDM4374g, and TDM4688g (Girish et al. 2012; Igawa et al. 2012). PK parameters for trastuzumab emtansine, total trastuzumab, and DM1 were consistent across the four studies at Cycle 1 and steady state. Trastuzumab emtansine PK was not affected by residual trastuzumab from prior therapy or circulating extracellular domain of HER2. No significant correlations were observed between

trastuzumab emtansine exposure and efficacy, thrombocytopenia, or increased concentrations of transaminases. Across the four studies, the incidence of anti-therapeutic antibodies to trastuzumab emtansine was low and detected in 4.5% (13/286) of evaluable patients receiving trastuzumab emtansine q3w.

The PK profile (i.e., maximum concentration  $[C_{max}]$ , area under the serum concentration-time curve [AUC], terminal half-life  $[T_{1/2}]$ , apparent volume of distribution at steady state  $[V_{ss}]$ , and CL) of single agent trastuzumab emtansine (3.6 mg/kg q3w) is predictable, well characterized, and unaffected by circulating levels of HER2 extracellular domain or residual trastuzumab. Trastuzumab emtansine exposure does not correlate with clinical responses or key AEs. Weekly administration of trastuzumab emtansine in study TDM3568g at a dose of 2.4 mg/kg showed consistent PK data with the q3w dosing schedule (Krop et al. 2008).

#### 1.2.2 CAPECITABINE

Capecitabine (Xeloda<sup>®</sup>) is a fluoropyrimidine carbamate with antineoplastic activity. It is an orally administered systemic prodrug of 5'-deoxy-5-fluorouridine (5'-DFUR) which is converted to 5-fluorouracil in the tumor, where it inhibits DNA synthesis and slows down tumor tissue growth. It has been evaluated in clinical trials in combination with docetaxel and as monotherapy in BC (Geyer et al. 2006; Wardley et al. 2006; von Minckwitz et al. 2011). Please see the national Xeloda<sup>®</sup> prescribing information or Investigator brochure for more information.

#### 1.2.2.1 Study BO18255: Capecitabine and Trastuzumab in mGC

Recently, a global phase III study (ToGA trial, BO18255) of trastuzumab plus chemotherapy as first-line treatment for advanced HER2-positive GC was conducted in 584 patients previously untreated for HER2-positive inoperable locally advanced or recurrent and/or metastatic adenocarcinoma of the stomach or GEJ. Patients received either capecitabine or fluorouracil combined with cisplatin or the same chemotherapy in combination with trastuzumab. The primary study endpoint was OS, defined as the time from the date of randomization to the date of death from any cause. At the time of the analysis a total of 349 randomized patients had died: 182/290 patients (62.8%) in the control arm and 167/294 patients (56.8%) in the treatment arm. The majority of the deaths were due to events related to the underlying cancer (Bang et al. 2010).

Most patients enrolled in the study were male (76%); 52.9% were Asian and 37.7% were white. The primary tumor site was the stomach for 81.8% of patients, with the others having GEJ tumors. The addition of trastuzumab to chemotherapy resulted in an increase in median OS from 11.1 months to 13.8 months (HR 0.74, p = 0.0046). Objective response rate (47% *versus* 35%), PFS (6.7 *versus* 5.5 months), and TTP (7.1 *versus* 5.6 months) were also significantly increased with the addition of trastuzumab to chemotherapy compared to chemotherapy alone.
With regard to OS, a treatment effect could not be excluded in any predefined subgroup, including primary tumor site, histologic subtype, method of determining HER2-positivity, performance status, chemotherapy regimen, age, gender, and region of enrollment. A multivariate analysis for OS showed a consistent result, with an adjusted HR of 0.72 (p = 0.0036); variables found to influence primary outcome included Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1 *versus* 2), prior gastrectomy, and Asian region of enrollment (data on file). A multivariate analysis of OS for patients enrolled in Japan, from which the bulk of Asian patients were enrolled, demonstrated a HR of 0.68. This was consistent with the overall study results (Sawaki et al. 2011).

A pre-planned subgroup analysis by IHC score indicated that positive treatment effects are greater in tumors with higher levels of HER2 expression. Among patients whose tumors had these higher levels of HER2 expression, the median OS was 11.8 months *versus* 16 months (HR 0.65; 95% CI 0.51–0.83) and median PFS was 5.5 months *versus* 7.6 months (HR 0.64; 95 % CI 0.51–0.79) for chemotherapy *versus* chemotherapy plus trastuzumab respectively. For OS, the HR was 0.75 (95% CI 0.51–1.11) in the IHC 2 + /FISH + group and 0.58 (95% CI 0.41–0.81) in the IHC 3+/FISH+ group (Bang et al. 2010).

The addition of trastuzumab to chemotherapy did not result in an increased incidence of severe (Grade 3–4) or fatal (Grade 5) AEs. There were no additional significant safety issues with trastuzumab used in the treatment of advanced GC over and above those observed when it was used to BC. Taken together, the results of the ToGA trial (BO18255) not only demonstrate the role of HER2 suppression in the treatment of HER2-positive GC but also show that HER2-directed therapies can be added to conventional chemotherapy regimens without substantial increases in toxic side effects.

# 1.2.3 PRECLINICAL DATA OF THE COMBINATION OF TRASTUZUMAB EMTANSINE AND A FLUOROPYRIMIDINE

In breast cancer preclinical models an additive anti-tumor activity was observed with combinations of trastuzumab emtansine and 5FU (see Figure 2, [Lewis Phillips et al. 2008]). In GC models a similar additive effect was observed with trastuzumab emtansine and capecitabine (see Figure 3, [data on file]).

Figure 2 MMTV HER2 Fo5 Mammary Tumor Transplants



T-DM1 = trastuzumab emtansine; 5-FU = 5-fluoruracil



Figure 3 Anti-tumor Activity of Trastuzumab Emtansine in Combination with Capecitabine in NCI-N87

T-DM1 = trastuzumab emtansine; 5-FU = 5-fluoruracil

# 1.3 STUDY RATIONALE AND BENEFIT-RISK ASSESSMENT

## 1.3.1 FOR MBC

At present, mBC remains an incurable disease. The primary goal of treatment is maximizing the patient's survival and quality of life.

HER2-positive breast tumors have shown to benefit from anti-HER2 therapy. Regimens using the combination of anti-HER2 agents and chemotherapy have demonstrated higher efficacy than single agent therapy. As a consequence several different combination therapies have been approved for HER2-positive mBC treatment in most countries and are considered the current standard of care.

The combination of capecitabine with anti-HER2 therapies has demonstrated to be beneficial for mBC patients. The combination of capecitabine and lapatinib is approved in the United States since March 2007 for the treatment of HER2-positive mBC patients who have previously received an anthracycline, a taxane, and trastuzumab. In June 2008, the European Commission granted conditional marketing authorization for lapatinib in combination with capecitabine for the treatment of HER2-positive advanced or mBC patients who have previously received and progressed on an anthracycline, a taxane, and trastuzumab in the metastatic setting. The combination of capecitabine and trastuzumab has demonstrated significant efficacy benefit when compared to capecitabine alone (von Minckwitz et al. 2011).

In study TDM4450g, trastuzumab emtansine as a single agent showed a significant increase in PFS compared to the current standard of care of trastuzumab and a taxane (see Section 1.2.1.4), together with a favorable safety profile.

The Phase III, TDM4370g trial met its co-primary endpoint of improving PFS (by IRC) compared to those who received the combination of lapatinib and capecitabine (see Section 1.2.1.6).

Based on the mentioned studies, the combination of trastuzumab emtansine and capecitabine could provide the potential for enhanced anti-tumor efficacy in mBC, compared to single agent trastuzumab emtansine or trastuzumab in combination with chemotherarapy.

Furthermore, preclinical data suggest that the combination of trastuzumab emtansine and capecitabine has an additive effect (see Section 1.2.3).

Approximately 2000 patients with breast cancer have been treated in trastuzumab emtansine clinical trials with an acceptable safety profile and a positive risk-benefit ratio. A safety monitoring is in place to avoid potential overlapping toxicities. A broad development program is in place to seek approval for indications for mBC. Capecitabine in combination with anti-HER2 agent is a proven efficacious regimen with a well established safety profile in mBC. Trastuzumab emtansine and capecitabine have no known significant overlapping toxicities. Therefore, exploring the benefit of combination therapy of trastzumab emtansine and capecitabine in mBC patients seems justified.

## 1.3.2 FOR MGC

As for mBC, the primary goal of treatment for metastatic gastric cancer (mGC) is the maximizing of the patient's survival and quality of life.

HER2-positive gastric tumors have shown to benefit from anti-HER2 therapy. Regimens using the combination of anti-HER2 agents and chemotherapy have demonstrated higher efficacy than single agent therapy. As a consequence several different combination therapies have been approved for HER2-positive mGC treatment in most countries and are considered the current standard of care.

In HER2-positive mGC, the ToGA study (BO18255) has proven that the combination of chemotherapy and trastuzumab significantly improves OS (see Section 1.2.2.1) in this population. Fluropyrimidine based therapies (capecitabine, 5-fluorouracil) are the standard of care in mGC in general and were also the most frequent combination agents used in the ToGA trial (BO18255) (see Section 3.3.2).

Furthermore, preclinical data suggest that the combination of trastuzumab emtansine and capecitabine has an additive effect (see Section 1.2.3).

A development program for trastuzumab emtansine is in place to seek approval for mGC indications. Capecitabine in combination with anti-HER2 agent is a proven efficacious regimen with a well established safety profile in mGC. Trastuzumab emtansine and capecitabine might have overlapping

toxicities and therefore a safety monitoring is in place to avoid exposing patients to harm. Therefore, exploring the benefit of combination therapy of trastzumab emtansine and capecitabine in mGC patients seems justified.

# 2. OBJECTIVES

# 2.1 PHASE I: MTD FINDING OF TRASTZUMAB EMTANSINE AND CAPECITABINE IN MBC

#### 2.1.1 PRIMARY OBJECTIVE

 To determine the MTD of the combination of trastuzumab emtansine and capecitabine in mBC patients

# 2.1.2 SECONDARY OBJECTIVES

- Pharmacokinetics of trastuzumab emtansine and metabolites and capecitabine
- Safety of the combination of trastuzumab emtansine and capecitabine
- Overall response rate (ORR)

# 2.2 PHASE II: EXPLORATION OF EFFICACY IN MBC PATIENTS

## 2.2.1 PRIMARY OBJECTIVE

ORR by investigator assessment

# 2.2.2 SECONDARY OBJECTIVES

- Safety profile of the combination at the dose established during Phase I
- Time to response (TTR)
- Duration of response (DoR)
- Time to progression (TTP)
- Time to treatment failure (TTF)
- Progression free survival (PFS)
- Clinical benefit rate (CBR)
- Overall survival (OS)

# 2.3 PHASE I: MTD FINDING OF TRASTZUMAB EMTANSINE AND CAPECITABINE IN MGC

#### 2.3.1 PRIMARY OBJECTIVE

 To determine the MTD of the combination of trastuzumab emtansine and capecitabine in mGC patients

## 2.3.2 SECONDARY OBJECTIVES

- Pharmacokinetics of trastuzumab emtansine and metabolites and capecitabine
- Safety of the combination of trastuzumab emtansine and capecitabine
- Overall response rate (ORR)

# 3. <u>STUDY DESIGN</u>

# 3.1 DESCRIPTION OF STUDY

This is an international, multicenter Phase I/II dose finding study of two dosing schedules of trastuzumab emtansine and capecitabine combination therapy in HER2-positive mBC and locally advanced or mGC patients. The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in a Phase I study in both mBC and locally advanced or mGC patients. The MTD will also be assessed for anti-tumor effects (exploration of efficacy) in a Phase II, single arm study in the mBC cohort. There will be no exploration of efficacy in the mGC cohort.

## 3.1.1 OVERVIEW OF STUDY DESIGN

# **Overview of Study Design**

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine, in HER2-positive mBC and locally advanced or mGC patients, using a Phase I design, followed by a Phase II single arm study to explore the efficacy of the combination in mBC patients. There will be no exploration of efficacy in the mGC cohort. Results from the Phase I in mGC will be used as supporting information for future studies in the indication.

Cohort 1 for mBC patients will open first and MTD will be established. Once MTD is established, both Phase II for mBC patients and Cohort 2 for mGC patients will open.

An overview of the study design is depicted in Figure 4.

# **Duration of Treatment and Patient Follow-up**

<u>Length of treatment:</u> All patients will be treated until disease progression, intolerable toxicity, withdrawal of consent, or death.

<u>Patient follow-up:</u> All patients from both cohorts will be followed up until intolerable toxicity, withdrawn consent, death or up to a maximum of 2 years after the last patient was enrolled in the Phase II part of the study, whichever occurs first.

# **Duration of Study, Data Base Closure and Data Reporting**

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to be 2 years for dose finding and the Phase II/ Exploration of Efficacy. The study will end after the follow-up period was completed, as defined above. Last patient last visit (LPLV) is defined as the

last data collection point that can be either a clinic visit or a lab sample. At that time point, the database will be closed.

In the case that in Cohort 1 the dose level 1 is too toxic (>1/3 or >1/6 of dose limiting toxicity [DLT]), the combination may be considered unfeasible. Enrollment will be closed and no other cohort will be opened. Patients, who at that point, experience response as per RECIST will be offered the possibility to continue on trastuzumab emtansine as a single agent.

Data may be reported at the end of each cohort i.e. once the MTD for Cohort 1 has been defined and the dose for Phase II/Exploration of Efficacy has been selected. The latest point to write the Clinical Study Report (CSR) will be one year after database closure.

# **Treatment of Patients after Database Closure**

If at the moment of study closure there are patients who have not progressed and are still receiving study treatment, they will be offered the possibility to continue treatment by enrolling in an extension study.

Figure 4 Overview of Study Design



<sup>&</sup>lt;sup>1</sup> Capecitabine doses are administered daily on days 1 to 14 of the 3-week cycles

mBC = metastatic breast cancer; mGC = metastatic gastric cancer; MTD = maximum tolerated dose; q3w = every 3 weeks; qw = weekly; T-DM1 = trastuzumab emtansine

A schedule of assessments is provided in Appendix 1.

<sup>&</sup>lt;sup>2</sup> The MTD defined in mBC Phase I will be implemented in mBC Phase II and mGC Phase I

<sup>&</sup>lt;sup>3</sup> Cohort 2 will open to recruit mGC patients once the MTD is defined in Phase I for mBC patients

<sup>&</sup>lt;sup>4</sup> Patients on MTD in Phase I must re-consent, recruitment will be extended to 110 mBC patients

# 3.1.1.1 Overview of Phase I Design in mBC Patients

An overview of the Phase I study design is depicted in **Figure 5**.

Figure 5 Overview of Phase I Dose Finding Study Design



<sup>&</sup>lt;sup>1</sup> If Dose level 1 is too toxic (>1/3 or >1/6 DLT), the study will be terminated. DLT = dose limiting toxicity; MTD = maximum tolerated dose

#### **Determination of the Maximum Tolerated Dose in mBC Patients**

The trial will first investigate the feasibility of the combination of capecitabine and trastuzumab emtansine q3w in one cohort up to 18 patients, by escalating the dose of capecitabine from 750 mg/m² bid to 1000 mg/m² bid on days 1 to 14 in cycles of 3 weeks with a 3 by 3 classical Phase I design. Cohort 1 will open first and enroll patients with HER2-positive mBC.

#### **Enrollment into Cohort 1**

# Dose finding in mBC patients (Phase I)

According to the 3 by 3 classical study design, Cohort 1 will start with the enrollment of 3 patients at dose level 1. Patients will be evaluated for DLTs as specified in DLT definition (see Section 5.1.4). The dose tested of trastuzumab emtansine will remain fixed at 3.6 mg/kg q3w and 3 dose levels of capecitabine administered bid on days 1 to 14 in 3-week cycles will be tested.

The following doses will be explored in Cohort 1:

- **Dose level 1:** 750 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine
- Dose level 2: 850 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine
- Dose level 3: 1000 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine

If dose level 1 is found to be too toxic (DLT >1/3 or >1/6), the enrollment will be closed and the study will be terminated. The following escalation rules will be applied during the dose finding treatment phase:

- Step 1: Three patients will be enrolled at dose level 1
- Step 2: The toxicity of dose level 1 will be monitored and the following actions taken:
  - a) If none of these three patients (0/3) experiences a DLT, escalation to dose level 2 will occur
  - b) If one of the initial three patients (1/3) experiences a DLT, an additional three patients should be enrolled and treated at the same dose, i.e. dose level 1
  - c) If no more patients experience a DLT (1/6), escalation to the next dose level will occur
  - d) If one or more patients experience a DLT (>1/6), the MTD will be established as the immediate inferior dose level or the study may be terminated if it happens at dose level 1.
- Step 3: Step 2 should be repeated until the MTD is reached
  If the last dose exceeds the MTD, de-escalation to the previous dose should occur. This dose should be defined as MTD if 6 or more patients

have been safely treated at this dose level and no more than 1/6 of the patients experienced a DLT at that dose level.

If only 3 patients have been treated at this dose level, then 3 more patients will be treated and observed at this level in order to achieve at least 6 patients treated at the same dose level.

In order to define the dose for the Phase II/exploration of efficacy part of the study, the Steering Committee will evaluate not only the DLTs during Cycle 1 but also all available safety information during the subsequent cycles. The dose level considered optimal by the Steering Committee will be the dose level selected to move forward with in the Phase II and mGC parts of the study.

Once the appropriate dose of study medication is established, the other cohorts will open as per Figure 4.

# 3.1.1.2 Overview of Phase II: Exploration of Efficacy in mBC Patients

Once the Steering Committee has defined the MTD to treat patients in Phase II, additional 90–100 mBC patients will be enrolled.

Only the mBC patients who have received the MTD dose from Phase I will continue with the Phase II part of the study to assess efficacy and safety of this treatment combination of capecitabine and trastuzumab emtansine.

See Section 3.1.1 for further information.

# 3.1.1.3 Overview of Phase I Design in mGC Patients

## **Determination of MTD in mGC patients**

Cohort 2 will open when the capecitabine MTD is established for Cohort 1 and enroll HER2-positive locally advanced and mGC patients. Trastuzumab emtansine will be administered qw at the fixed dose of 2.4 mg/kg and capecitabine will be started at the MTD defined for mBC patients in Cohort 1. See Section 3.1.1 for further information.

# **Enrollment into Cohort 2**

Cohort 2 will open with a 3 by 3 classical design to investigate the feasibility of combination therapy of capecitabine and trastuzumab emtansine in Cohort 2 (enrolling up to 18 mGC patients) by escalating or de-escalating the dose of capecitabine starting from the MTD determined in Cohort 1. In case the MTD was not established or the enrollment was stopped for Cohort 1, enrollment into Cohort 2 will not take place.

The dose levels for escalation or de-escalation of capecitabine will be the same as described for Cohort 1:

- a) If the MTD in Cohort 1 was defined at dose level 1 of 750 mg/m<sup>2</sup> bid
  - If dose level 1 is tolerated, doses should be escalated to dose level 2 of 850 mg/m² bid

- If dose level 1 is not tolerated (>1/3 or >1/6 DLT), the combination will be considered not feasible and Cohort 2 will be terminated
- b) If the MTD in Cohort 1 was defined at dose level 2 of 850 mg/m<sup>2</sup> bid
  - If dose level 2 is tolerated, doses should be escalated to dose level 3 of 1000 mg/m² bid
  - If dose level 2 is not tolerated, doses should be de-escalated to dose level 1 of 750 mg/m² bid
- c) If the MTD in Cohort 1 was defined at dose level 3 of 1000 mg/m<sup>2</sup> bid
  - olf dose level 3 is tolerated, no escalation will be done and the MTD will be defined at dose level 3
  - olf dose level 3 is not tolerated, doses should be de-escalated to dose level 2 of 850 mg/m² bid

# 3.1.1.4 Considerations for all Patients Treated in the Study

Safety data will be reviewed on an ongoing basis (i.e. real time safety monitoring) by the Steering Committee. The preliminary safety review will be based on the safety information (DLTs, dose delays, dose reductions and Grade 3–5 events) observed during the first cycle in at least 3 patients.

#### 3.1.1.5 Number of Patients

Overall, it is anticipated that the maximum number of patients enrolled into the study will be 140 patients.

#### Phase I: mBC

From 3–18 patients will be enrolled into Cohort 1 to determine the MTD of capecitabine in combination with trastuzumab emtansine in mBC patients.

# Phase II: Exploration of Efficacy in mBC

For this part of the study, Cohort 1 will be expanded to 110 mBC patients.

## Phase I: mGC

After the MTD in Cohort 1 has been established, 3–18 patients will be enrolled into Cohort 2 to determine the MTD of capecitabine in combination with trastuzumab emtansine in mGC patients.

## 3.1.1.6 Number of Centers

This is a multicenter, international study.

## 3.1.2 STEERING COMMITTEE

A Steering Committee has been established for this study. Initially, it is composed of the investigators participating in the Phase I Cohort 1 part of the study and one medical representative and one statistician of the Sponsor. The study design and DLT has been developed by the Steering Committee. See Steering Committee Charter for further information.

End of study is defined as LPLV at the end of the follow-up period as defined in Section 3.1.1.

## 3.3 RATIONALE FOR STUDY DESIGN

#### 3.3.1 RATIONALE FOR PATIENT GROUP SELECTION

Nonclinical studies indicate that the sensitivity of cancer cells to trastuzumab emtansine requires HER2 overexpression, and measurement of such expression is a standard of care in determining eligibility for trastuzumab therapy (see the Herceptin<sup>®</sup> national prescribing information). Measurement of HER2 gene amplification has traditionally been performed using IHC measurement. HER2 gene amplification determined by FISH has also proven to be a reliable method for demonstrating HER2-positive status (Press et al. 2005).

This study will enroll patients diagnosed with the disease to which the combination is intended. The combination of anti-HER2 agent and capecitabine has shown to be efficacious in both mBC (von Minckwitz et al. 2011; Geyer et al. 2006) and mGC (Bang et al. 2010), and capecitabine is a standard of care treatment for both diseases. Both diseases have been shown to benefit from anti-HER2 treatment; therefore, all patients must be diagnosed with HER2-positive disease. Patients with incurable mBC and locally advanced or mGC whose tumors are positive for HER2 overexpression represent the patient population eligible for study enrollment.

# 3.3.1.1 Rationale for Phase I

The study design of 3 by 3 Phase I is well established and well known method for Phase I studies. PK parameters will be collected and analyzed in order to investigate the PK interaction of the drugs under investigation. Since both agents are administered at efficacious doses, the risk of enrolling patients at the sub-optimal doses is minimal.

## 3.3.1.2 Rationale for Phase II

Phase II is designed to provide an estimation of the treatment effect of the combination at the selected MTD. In addition, it will provide important information on the longer term safety of the combination.

# 3.3.2 RATIONALE FOR INVESTIGATIONAL MEDICINAL DOSE SELECTION

#### 3.3.2.1 In mBC Patients

In study TDM3569g, the MTD of trastuzumab emtansine administered by IV infusion q3w was 3.6 mg/kg. As described in Section 1.2, clinical activity has been observed at a dose of 3.6 mg/kg q3w in two Phase II studies of single-agent trastuzumab emtansine in patients with advanced heavily pre-treated HER2-positive mBC (protocol TDM4258g and protocol TDM4374g)

and in patients who had not received prior chemotherapy for metastatic disease (TDM4450g).

Capecitabine doses have been selected as being in the range of efficacious doses for single agent or combination use. The dose of 750 mg/m² bid was considered the minimum efficacious dose. The maximum dose of 1000 mg/m² bid is the currently approved dose of capecitabine (please see the current national prescribing information of Xeloda®).

#### 3.3.2.2 In mGC Patients

In the ToGA study (BO18255: trastuzumab in combination with chemotherapy in mGC), patients with higher drug exposure had a greater benefit compared to those with lower exposure (Yang et al. 2011). As a consequence, a randomized, open label, multicenter Phase IIIb study comparing two trastuzumab dosing regimens, each in combination with cisplatin/capecitabine chemotherapy, as first line therapy in patients with HER2-positive metastatic gastric or gastro-esophageal junction adenocarcinoma is being conducted (Study BO27798).

In TDM3569g (see Section 1.2.1.1), the qw administration of 2.4 mg/kg of trastuzumab emtansine resulted in higher exposure (see Section 1.2.1.7) (Krop et al. 2008). Therefore, this dose may result in larger clinical benefit for mGC patients. Trastuzumab emtansine at 2.4 mg/kg qw is being tested in the BO27952 study.

In Cohort 2, the starting dose of capecitabine will be the MTD from Cohort 1 (mBC) in order to minimize the exposure of patients to sub-optimal treatment. The dose of capectiabine can be de-escalated if needed.

# 3.3.2.3 Rationale for Duration of Treatment

Treatment will be given until disease progression or unacceptable toxicity (see Section 3.1.1 for full information). As of 1 January 2010, of 237 patients enrolled in studies TDM3569g, TDM4258g, and TDM4374g receiving trastuzumab emtansine at 3.6 mg/kg, approximately 30% have tolerated more than 12 cycles, with 14.8% having received more than 17 cycles. Twenty patients (8.4%) have discontinued trastuzumab emtansine due to AEs and 24 patients (10.1%) required dose reductions in trastuzumab emtansine because of AEs. In the absence of intolerable toxicity, patients with mBC are generally treated until disease progression.

Capecitabine will be given until disease progression, as per Xeloda<sup>®</sup> national prescribing information.

## 3.3.3 PHARMACOKINETIC SAMPLING RATIONALE

The PK sampling rationale is to characterize the pharmacokinetics of trastuzumab emtansine, total trastuzumab, and DM1, to assess potential drug-drug interaction when trastuzumab emtansine is given in combination with capecitabine, and to explore potential correlations between drug exposure and measures of both efficacy (ORR) and toxicity (ALT/AST, platelets, etc.), if data allow.

## 3.4 OUTCOME MEASURES

# 3.4.1 PHASE I: MBC

# 3.4.1.1 Primary Efficacy Outcome Measure

The main objective for Phase I is to determine the MTD of capecitabine when combined with trastuzumab emtansine.

# 3.4.1.2 Secondary Efficacy Outcome Measure

The secondary outcome is ORR, based on best overall response rate (BORR) as per RECIST v.1.1; based on investigator assessment.

# 3.4.1.3 Primary Safety Outcome Measure

The primary outcome measure is to establish MTD.

# 3.4.1.4 Secondary Safety Outcome Measures

Safety endpoints will be summarized for both treatment phases: dose finding and exploration of efficacy. Again, the summary of safety endpoints will be presented for each cohort:

- Incidence, nature and severity of AEs, as per NCI CTCAE v. 4.0
- Incidence, nature, and severity of serious AEs
- Incidence and nature of AEs equal or higher than Grade 3
- Premature withdrawal from study and study medication
- Abnormal laboratory values
- LVEF
- Exposure to study medication
- Concomitant medications and physical examination

#### 3.4.1.5 Pharmacokinetic Outcome Measures

The PK outcome measures to be assessed in patients receiving trastuzumab emtansine and capecitabine will include:

- Serum concentrations of trastuzumab emtansine (conjugated drug) and total trastuzumab (free and conjugated to DM1)
- Plasma concentration of DM1
- Plasma concentration of capecitabine and its active metabolite 5fluorouracil (5-FU)

## 3.4.2 Phase II: Exploration of Efficacy: MBC

# 3.4.2.1 Primary Efficacy Outcome Measure

The primary outcome measure is ORR, based on best overall response (BOR) (defined as the best response recorded from the start of treatment until

disease progression/recurrence or death; or for newly enrolled patients the best response from the start of Phase II until disease progression or death) by investigator assessment; as per RECIST v.1.1 Appendix 3.

# 3.4.2.2 Secondary Efficacy Outcome Measures

Secondary outcomes include:

- Time to response (TTR)
- Duration of response (DoR)
- Time to progression (TTP)
- Time to treatment failure (TTF)
- Progression free survival (PFS)
- Clinical benefit rate (CBR)
- Overall survival (OS)

# 3.4.2.3 Primary Safety Outcome Measure

A primary safety outcome is defined only for Phase I.

# 3.4.2.4 Secondary Safety Outcome Measures

Safety endpoints will be summarized for both treatment phases: dose finding and exploration of efficacy. Again, the summary of safety endpoints will be presented for each cohort:

- Incidence, nature and severity of AEs, as per NCI CTCAE v. 4.0
- Incidence, nature, and severity of serious AEs
- Incidence and nature of AEs equal or higher than Grade 3
- Premature withdrawal from study and study medication
- Abnormal laboratory values
- LVEF
- Exposure to study medication
- Concomitant medications and physical examination

## 3.4.2.5 Pharmacokinetic Outcome Measures

Not applicable for Phase II.

# 3.4.3 Phase I: MGC

# 3.4.3.1 Primary Efficacy Outcome Measure

The main objective for Phase I is to determine the MTD of capecitabine when combined with trastuzumab emtansine.

# 3.4.3.2 Secondary Efficacy Outcome Measure

The secondary outcome is ORR, based on BORR as per RECIST v.1.1; based on investigator assessment.

# 3.4.3.3 Primary Safety Outcome Measure

The primary outcome measure is to establish MTD

# 3.4.3.4 Secondary Safety Outcome Measures

Safety endpoints will be summarized for both treatment phases: dose finding and exploration of efficacy. Again, the summary of safety endpoints will be presented for each cohort:

- Incidence, nature and severity of AEs, as per NCI CTCAE v. 4.0
- Incidence, nature, and severity of serious AEs
- Incidence and nature of AEs equal or higher than Grade 3
- Premature withdrawal from study and study medication
- Abnormal laboratory values
- LVEF
- Exposure to study medication
- Concomitant medications and physical examination

## 3.4.3.5 Pharmacokinetic Outcome Measures

The PK outcome measures to be assessed in patients receiving trastuzumab emtansine and capecitabine will include:

- Serum concentrations of trastuzumab emtansine (conjugated drug) and total trastuzumab (free and conjugated to DM1)
- Plasma concentration of DM1
- Plasma concentration of capecitabine and its active metabolite 5fluorouracil (5-FU)

# 4. MATERIALS AND METHODS

# 4.1 PATIENTS

# 4.1.1 MBC PATIENTS

This study will enroll HER2-positive BC patients with histologically or cytologically confirmed metastatic disease which are amenable for combination treatment with trastuzumab emtansine and capecitabine.

Metastatic BC patients must have received at least one treatment regimen which includes a chemotherapy and trastuzumab agent. Only patients whose HER2 tumor status was locally scored as IHC 3+ or ISH positive will be permitted for both study parts (Phase I and II).

## 4.1.2 MGC PATIENTS

This study will enroll HER2-positive GC patients with histologically or cytologically confirmed inoperable locally advanced or metastatic disease which are amendable for combination treatment with trastuzumab emtansine and capecitabine.

Metastatic GC patients must have not received prior chemotherapy for advanced/metastatic disease, and only patients with HER2-positive primary tumor or metastasis as assessed by central laboratory will be allowed to enroll in dose finding part for this disease in this study.

## 4.1.3 INCLUSION CRITERIA

#### 4.1.3.1 For mBC Patients

Patients must meet the following criteria for study entry:

- 1. Age ≥ 18 years old
- 2. Signed informed consent prior to any study specific procedure
- 3. Able and willing to comply with protocol
- 4. Negative serum pregnancy test for women of childbearing potential (including pre menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential
- 5. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 6 months after the last dose of study treatment (see Section 5.2.4)
- 6. ECOG performance status of 0, 1, or 2
- 7. Blood:
  - a) Platelet count > 100,000 cells/mm<sup>3</sup>
  - b) International normalized ratio (INR) < 1.5 × the upper limit of normal (ULN)</li>
  - c) Absolute neutrophil count (ANC) > 1500 cells/mm<sup>3</sup>
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 8. Liver function:
  - a) Total bilirubin ≤ 1.5 × ULN except in patients with previously documented Gilbert's syndrome in which case total bilirubin ≤ 3 mg/dL is acceptable

- b) Serum glutamic oxaloacetic transaminase (SGOT)/AST and serum glutamic pyruvic transaminase (SGPT)/alanine transaminase (ALT) ≤ 2.5 × the ULN
- c) Alkaline phosphatase ≤ 2.5 × the ULN. Patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × the ULN
- 9. Renal function:
  - a) Serum creatinine of < 177 µmol/L or calculated creatinine CL > 50 mL/min. I urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24 hour urine collection and demonstrate ≤ 1 g of protein/24 hours
- 10. Cardiac function:
  - a) LVEF ≥ 50% by echocardiogram (ECHO) or multiple-gated acquisition (scan) (MUGA)
- 11. Histologically or cytologically confirmed breast cancer
- 12. HER2-positive disease IHC 3+ or ISH positive
- 13. Tumor block available or 15 slides for retrospective central confirmation of HER2-positivity (central confirmation not necessary for enrolment)
- 14. Metastatic breast cancer (mBC) with at least one measurable lesion according to RECIST
- 15. Disease progression on at least one regimen containing trastuzumab and chemotherapy
- 16. Patients must have recovered from previous treatments

#### 4.1.3.2 For mGC Patients:

Patients must meet the following criteria for study entry:

- 1. Age ≥ 18 years old
- 2. Signed informed consent prior to any study specific procedure
- 3. Able and willing to comply with protocol
- 4. Negative serum pregnancy test for women of childbearing potential (including pre menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential
- 5. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 6 months after the last dose of study treatment (see Section 5.2.4)
- 6. ECOG performance status of 0, 1, or 2
- 7. Blood:

- a) Platelet count > 100,000 cells/mm<sup>3</sup>
  - b) INR  $< 1.5 \times$  the ULN
  - c) ANC > 1500 cells/mm<sup>3</sup>
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 8. Liver function:
  - a) Total bilirubin ≤ 1.5 × ULN except in patients with previously documented Gilbert's syndrome in which case total bilirubin ≤ 3 mg/dL is acceptable
  - b) SGOT/AST and serum glutamic pyruvic transaminase (SGPT)/ALT ≤ 2.5 × the ULN
  - c) Alkaline phosphatase ≤ 2.5 × the ULN. Patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × the ULN
- 9. Renal function:
  - a) Serum creatinine of < 177 μmol/L or calculated creatinine CL > 50 mL/min. I urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24 hour urine collection and demonstrate ≤ 1 g of protein/24 hours
- 10. Cardiac function:
  - a) LVEF ≥ 50% by ECHO or MUGA
- 11. Histologically or cytologically confirmed GC
- 12. HER2-positive tumor (primary tumor or metastatic lesion), defined as either IHC 3+ alone or IHC 2+ in combination with ISH+, prospectively confirmed by a Sponsor-designated central laboratory prior to enrollment. ISH positivity is defined as a ratio of ≥ 2.0 for the number of HER2 gene copies to the number of signals for CEP17.
  - a) Archival tumor samples obtained from primary or metastatic sites are acceptable.
  - b) Invasive tumor for central confirmation of HER2 status is required.
  - c) A formalin-fixed paraffin-embedded (FFPE) tissue block with at least 5 mm of invasive tumor for central confirmation is preferred.
    - If FFPE tissue blocks (or partial block) are unavailable due to country or site regulations, a minimum of 8 freshly cut unstained slides MUST be available for central review of HER2 status.
- 13. Inoperable locally advanced or mGC

#### 4.1.4 EXCLUSION CRITERIA

## 4.1.4.1 For mBC Patients:

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half lives, whatever is longest

- c) Trastuzumab within 21 days
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received prior trastuzumab emtansine
- 3. Prior treatment with capecitabine
- 4. History of severe and unexpected reactions to fluoropyrimidine or with known hypersensitivity to fluorouracil
- 5. Related capecitabine contraindications:
  - a)Treatment with sorivudine or its chemically related analogues, such as brivudine
  - b)Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 360 mg/m<sup>2</sup>
  - b) Epirubicin > 900 mg/m<sup>2</sup>
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 360 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 28 days of first study drug administration
- 9. Current peripheral neuropathy of Grade ≥ 3 per the NCI CTCAE, v4.0
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above
- 11. Current unstable ventricular arrhythmia requiring treatment
- 12. History of symptomatic CHF (New York Heart Association [NYHA] Classes II–IV)
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
- 15. Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)

- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation
- 20. Current known active infection with human influenca virus (HIV), hepatitis B, and/or hepatitis C virus
  - a) For patients who are known carriers of hepatitis B virus (HBV), active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Lapatinib ≤ 14 days before first study drug administration
- 22. Previous radiotherapy for the treatment of unresectable, locally advanced/recurrent or mBC is not allowed if:
  - a) The last fraction of radiotherapy has been administered within 14 days prior to first study drug administration.
  - b) More than 25% of marrow-bearing bone has been irradiated.
  - c) The patient has not recovered from any resulting acute toxicity to Grade ≤ 1 prior to first study drug administration.

## 4.1.4.2 For mGC Patients:

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half lives, whatever is longest
  - b) Hormonal therapy within 14 days
  - c) Trastuzumab within 21 days
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received prior trastuzumab emtansine
- 3. Prior treatment with capecitabine
- 4. History of severe and unexpected reactions to fluoropyrimidine or with known hypersensitivity to fluorouracil
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically related analogues, such as brivudine
  - b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 360 mg/m<sup>2</sup>
  - b) Epirubicin > 900 mg/m<sup>2</sup>
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>

- d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 360 mg/m<sup>2</sup> doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 28 days of first study drug administration
- 9. Current peripheral neuropathy of Grade ≥ 3 per the NCI CTCAE, v4.0
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above
- 11. Current unstable ventricular arrhythmia requiring treatment
- 12. History of symptomatic CHF (New York Heart Association [NYHA] Classes II–IV)
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
- 15. Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation
- 20. Current known active infection with HIV, hepatitis B, and/or hepatitis C virus
  - a) For patients who are known carriers of hepatitis B virus (HBV), active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Previous chemotherapy for advanced/metastatic disease
  - a) Prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study

## 4.2 STUDY TREATMENT

# 4.2.1 FORMULATION, PACKAGING, AND HANDLING

## 4.2.1.1 Trastuzumab Emtansine

Trastuzumab emtansine is provided as a single-use, lyophilized formulation in a colorless 20 mL Type I glass vial containing 160 mg of trastuzumab emtansine, closed by means of a FluroTec coated stopper and an overseal with flip-off cap. Upon receipt of trastuzumab emtansine, vials should be refrigerated at 2–8°C (36–46°F) until use. THE VIAL MUST NOT BE FROZEN OR SHAKEN. Trastuzumab emtansine must be stored in the original carton to protect it from light. Do not use the product beyond the expiration date provided by the manufacturer. The reconstituted product contains no preservative and is intended for single use only. Any remaining medication should be discarded.

All vials of trastuzumab emtansine should be handled by appropriately trained site staff wearing gloves and using appropriate procedures in place at the clinical site for preparation of chemotherapeutic drugs. Vials should be visually inspected upon receipt to ensure that they are intact without exterior contamination. Discard any cracked vials and report vials with surface contamination to the clinical site manager for assessment.

The lyophilized product should be reconstituted using Sterile Water for Injection (SWFI). Using a new syringe, 8 mL SWFI should be added to the vial and the vial swirled gently until the product is completely dissolved. The vial should not be shaken. The resulting product contains 20 mg/mL trastuzumab emtansine, 10 mM sodium succinate, pH 5.0, 60 mg/mL sucrose, and 0.02% (w/v) polysorbate 20. Each 20 mL vial contains enough trastuzumab emtansine to allow delivery of 160 mg trastuzumab emtansine. The reconstituted product contains no preservative and is intended for single use only.

The vial should be inspected to ensure the reconstituted product is a clear colorless solution, and is free of particulates before proceeding. Drug from any vial that appears abnormal upon inspection should not be administered to patients. Using a new syringe, the indicated volume of trastuzumab emtansine solution should be removed from the vial(s) and added to the IV bag containing at least 250 mL of 0.45% sodium chloride (preferred) or 0.9% sodium chloride injection and gently inverted to mix the solution. A 0.22 micron non-protein adsorptive polyethersulfone in line filter is recommended when using 0.45% sodium chloride and required when using 0.9% sodium chloride injection. The solution of trastuzumab emtansine should not be shaken.

The solution of trastuzumab emtansine for infusion should be used immediately. If not used immediately, storage times should not be longer than 24 hours at 2–8°C (36–46°F) for solutions of trastuzumab emtansine diluted in polyvinyl chloride (PVC) or latex free PVC-free polyolefin, polypropylene, or polyethylene bags containing 0.45% or 0.9% Sodium Chloride for Injection.

Study MO28230

For additional details, please refer to the current version of the trastuzumab emtansine Investigator's Brochure.

# 4.2.1.2 Capecitabine

The following information has been obtained from the Xeloda<sup>®</sup> EU Summary of Product Characteristics and U.S. Xeloda<sup>®</sup> Package Insert.

Capecitabine is available as biconvex, oblong, film-coated tablets, available as follows:

- 150 mg tablets: color, light peach; engraving, XELODA on one side, 150 on the other; packs of 60
- 500 mg tablets: color, peach; engraving, XELODA on one side, 500 on the other; packs of 120

Capecitabine tablets should not be stored above 30°C.

# 4.2.2 DOSAGE AND ADMINISTRATION

## 4.2.2.1 For mBC Patients

#### Trastuzumab Emtansine

Trastuzumab emtansine will be administered on Day 1 of a 3-week cycle q3w at a dose of 3.6 mg/kg IV (see Appendix 1). The total dose will be calculated based on the patients weight on Day 1 (or up to 3 days before) of each cycle with no upper limit.

If the timing of trastuzumab emtansine coincides with a holiday that precludes the procedure, the procedure should be performed within 3 business days of the scheduled date and, when possible, on the earliest following date, with subsequent protocol-specified procedures rescheduled accordingly.

The first infusion of trastuzumab emtansine will be administered over 90 minutes (±10 minutes). Infusions may be slowed or interrupted for patients experiencing infusion associated symptoms. Vital signs must be assessed before and after dose administration. Following the initial dose, patients will be observed for at least 60 minutes for fever, chills, or other infusion associated symptoms. If prior infusions were well tolerated (without any signs or symptoms of infusion reactions), subsequent doses of trastuzumab emtansine may be administered over 30 minutes (±10 minutes), with a minimum 30 minute observation period following infusion. Local health authority guidelines must be followed with regard to further observation and monitoring, if applicable.

Pre-medication for nausea and infusion reactions (e.g., acetaminophen or other analgesics, antihistamines such as diphenhydramine, or corticosteroids) may be given at the investigator's discretion.

# Capecitabine

Capecitabine will be administered twice a day, orally for 14 days followed by a 7-day rest period at the dose levels 1–3 described in the "study design"

Section 3.1.1. Capecitabine tablets should be swallowed with water within 30 minutes after a meal.

If a dose is missed, the patient should skip that dose. The patient should not double the dose during the next administration.

For Phase II, guidelines for dosage modification and treatment interruption or discontinuation are provided in Section 5.1. For this part of the study, the MTD from Phase I will be used as a starting dose.

## 4.2.2.2 For mGC Patients

#### **Trastuzumab Emtansine**

Trastuzumab emtansine will be administered on Day 1 of a qw cycle qw at a dose of 2.4 mg/kg IV (see Appendix 1). The total dose will be calculated based on the patients weight on Day 1 (or up to 3 days before) of each cycle with no upper limit.

Administration time and observation period will be performed as described in Section 4.2.2.1 for trastuzumab emtansine.

Guidelines regarding timing delays and infusion times are the same as for mBC patients, as is the accepted pre-medication.

# Capecitabine

Capecitabine will be administered twice a day, orally, for 14 days followed by a 7-day rest period at the dose level that was determined during the dose finding part of the study in mBC patients as the MTD in Cohort 1. Capecitabine tablets should be swallowed with water within 30 minutes after a meal.

If a dose is missed, the patient should skip that dose. The patient should not double the dose the next administration.

Guidelines for dosage modification and treatment interruption or discontinuation are provided in Section 5.1.

## 4.2.3 Investigational Medicinal Product Accountability

All investigational medicinal products (IMPs) required for completion of this study (trastuzumab emtansine and capecitabine) will be provided by the Sponsor. The investigational site will acknowledge receipt of IMPs, using the interactive voice/web recognition system (IxRS) to confirm the shipment condition and content. Any damaged shipments will be replaced.

IMPs will either be disposed of at the study site according to the study site's institutional standard operating procedure or returned to the Sponsor with the appropriate documentation. The site's method of IMP destruction must be agreed upon by the Sponsor. The site must obtain written authorization from the Sponsor before any IMP is destroyed, and IMP destruction must be documented on the appropriate form.

Accurate records of all IMPs received at, dispensed from, returned to, and disposed of by the study site should be recorded on the Drug Inventory Log.

# 4.2.4 POST-TRIAL ACCESS TO EXTENSION STUDY

Post-trial access of trastuzumab emtansine and capecitabine will be performed as described in Section 3.1.1, *Treatment of Patients and Database Closure*. In case a patient decides to withdraw from the study, no post-trial access will be granted. Currently, the Sponsor does not have any plans to provide other study interventions to patients after conclusion of the study or any earlier patient withdrawal.

# 4.3 CONCOMITANT AND EXCLUDED THERAPIES

#### 4.3.1 PERMITTED THERAPY

Concomitant therapy and pre-medication are defined as non-IMPs.

Concomitant therapy includes any prescription medication, over-the-counter preparation, or herbal therapy between the 14 days preceding first treatment and the Study Treatment Discontinuation Visit. Afterwards, only anti-cancer therapies will be collected as part of the survival follow-up period.

Pre-medication is allowed according to standard practice guidelines.

No pre-medication for the first infusion of trastuzumab emtansine is required; however, pre-medication is allowed at the investigator's discretion.

Concomitant use of erythropoiesis stimulating agents is allowed if clinically indicated in accordance with local prescribing guidelines.

Palliative radiotherapy may be permitted to treat pre-existing painful bone metastases or to treat brain metastases (for patients who have disease control outside of the brain). Please contact the Medical Monitor for approval. If the Medical Monitor cannot be reached because of time zone differences, radiotherapy may be administered, but the Medical Monitor should still be informed.

Other medications considered necessary for the patient's safety and well being may be given at the discretion of the investigator. Use of bisphosphonates or denosumab is permitted for the control of bone pain, prevention and/or treatment of bony metastases, and treatment of osteoporosis. If bisphosphonates are required for the treatment of symptomatic malignancy-associated hypercalcemia, tumor assessments should be performed to assess for potential disease progression.

## 4.3.2 PROHIBITED THERAPY

Use of the therapies described below is prohibited during the study prior to discontinuation of study treatment (collectively, these will be referred to as non-protocol therapy).

Any therapies intended for the treatment of cancer, other than trastuzumab emtansine, whether they are approved by national health authorities or

experimental, including cytotoxic chemotherapy, immunotherapy, hormonal therapy (other than megestrol acetate), and biologic or targeted agents (other than granulocyte colony-stimulating factor and erythropoiesis stimulating agents), are prohibited.

Radiotherapy for unequivocal disease progression is not permitted while on study treatment, with the exception of new brain metastases or isolated progression of previously treated brain lesions. Patients who have disease control outside of the brain, defined as continued PR or CR of any duration, or SD for ≥3 months, but who have developed brain metastases that are treatable with radiation will be allowed to continue to receive study therapy until they either experience systemic progression of their disease and/or further progression in the brain that cannot be treated with additional radiation. Patients must not miss more than one cycle of study treatment for the treatment of their brain metastases and must have an ECOG performance status of 0, 1 or 2 to continue on therapy. The Medical Monitor should be informed before a decision is made to resume study treatment after radiotherapy for brain metastases.

## 4.4 STUDY ASSESSMENTS

All patients will be closely monitored for safety and tolerability during all cycles of therapy and at the safety follow-up visit:

- Visits will be based on a q3w cycle for mBC
- Visits will be based on a qw cycle for mGC

Study assessments are outlined in this section and in Appendix 1.

# 4.4.1 DESCRIPTION OF STUDY ASSESSMENTS

All patients will be closely monitored for safety and tolerability during all cycles of therapy and at the Study Treatment Discontinuation Visit. Patients should be assessed for toxicity prior to each dose; dosing will occur only if the clinical assessment and local laboratory test values are acceptable. Trastuzumab emtansine will be administered either in q3w cycles (mBC patients) or qw cycles (mGC patients) if no additional time is required for reversal of toxicity. Dose delays and dose reductions will be allowed for trastuzumab emtansine as outlined in Section 5.1.5.

If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend that precludes the procedure within the allotted window, the procedure should be performed on the nearest following date (i.e. within 3 business days).

# 4.4.1.1 Medical History and Demographic Data

Medical history includes clinically significant diseases, surgeries, cancer history (including prior cancer therapies and procedures), smoking history, use of alcohol and drugs of abuse, and all medications (e.g., prescription drugs, over-the-counter drugs, herbal/homeopathic remedies, nutritional supplements) used by the patient within 14 days prior to the screening visit.

Demographic data will include age, sex, and self-reported race/ethnicity.

# 4.4.1.2 Vital Signs

Vital signs will include measurements of weight, respiratory rate, heart rate, blood pressure, and temperature. Abnormal or significant changes to vital signs from baseline should be recorded as AEs, if appropriate.

# 4.4.1.3 Physical Examinations

A complete physical examination should include the evaluation of head, eye, ear, nose, and throat; cardiovascular; dermatological; musculoskeletal; respiratory; gastrointestinal; and neurological systems. Changes from baseline abnormalities should be recorded at each subsequent physical examination. New or worsened abnormalities should be recorded as AEs if appropriate.

As part of tumor assessment, physical examinations should also include the evaluation of the presence and degree of enlarged lymph nodes, hepatomegaly, and splenomegaly.

Limited physical examinations will be symptom-directed.

# 4.4.1.4 Tumor and Response Evaluations

Measurable and unmeasurable disease must be documented at screening and re-assessed at each subsequent tumor evaluation. Tumor assessments with computed tomography (CT) or magnetic resonance imaging (MRI) scans of the chest, abdomen, and pelvis are to be performed as described in Appendix 1, Schedule of Assessment. CT or MRI of the brain and baseline radioisotope bone scan must be obtained at screening. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to first treatment the bone scan does not need to be repeated and non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Tumor assessments should include an evaluation of all known and/or suspected sites of disease, whenever possible. Patients should have lesions selected that can be evaluated at every tumor assessment. The same radiographic procedure used at screening must be used throughout the study (e.g., the same contrast protocol for CT scans). Response assessments will be assessed by the investigator, based on physical examinations, CT or MRI scans, and bone scans using RECIST v. 1.1 (see Appendix 3). In the event a positron emission tomography (PET)/CT scanner is used for tumor assessments, the CT portion of the PET/CT must meet criteria for diagnostic quality. Please consult the Imaging Manual for guidelines on performing a diagnostic guality (optimized) CT exam. For patients who continue study treatment after isolated brain progression, the frequency of follow-up scans is at the discretion of the investigator.

At the investigator's discretion, CT scans, MRI scans, and/or bone scans may be obtained at any time when clinically indicated or if PD is suspected. If a bone scan cannot be performed during the course of the study because of the unavailability of the Tc-99m isotope, the investigator may choose an alternative imaging modality (see Appendix 4).

Radiographic imaging should always be performed rather than clinical examination unless the lesion(s) being followed cannot be imaged but are assessable by clinical examination. In applying RECIST, documentation by color photography including a ruler to estimate the size of the lesion is recommended

# 4.4.1.5 Laboratory Assessments

## For mBC Patients:

# **Local Laboratory Assessments:**

- Hematology, biochemistry, coagulation, urinalysis, and pregnancy testing
- Prospective HER2 status. Patients will be enrolled based on local results

# **Central Laboratory Assessments:**

- Retrospective HER2 status
- PK assays:
- Serum trastuzumab emtansine concentration and total trastuzumab using a validated immunoassay
- Serum capeciatbine and 5 follow-up PK samples
- Plasma concentration of DM1 using a validated liquid chromatography electrospray tandem mass spectrometry (LC-MS/MS) method

# For mGC Patients:

# **Local Laboratory Assessments:**

Hematology, biochemistry, coagulation, urinalysis, and pregnancy testing

# **Central Laboratory Assessments:**

- Prospective HER2 status. Patients will be enrolled based on central results
- PK assays:
- Serum trastuzumab emtansine concentration and total trastuzumab using a validated immunoassay
- Serum capeciatbine and 5 follow-up PK samples
- Plasma concentration of DM1 using a validated liquid chromatography electrospray tandem mass spectrometry (LC-MS/MS) method

# 4.4.1.6 Electrocardiograms

A 12-lead ECG should be obtained at baseline and be printed and kept with the patient's record.

#### 4.4.1.7 ECHO/MUGA

ECHO is the preferred modality because of the global technetium (Tc-99m) shortage (see Appendix 4). The same method used at screening should be used throughout the study.

## 4.4.2 TIMING OF STUDY ASSESSMENTS

# 4.4.2.1 Screening and Pretreatment Assessments

Written informed consent for participation in the study must be obtained before performing any study specific screening tests or evaluations. Informed Consent Forms for enrolled patients and for patients who are not subsequently enrolled will be maintained at the study site.

Once the patient has signed the Informed Consent Form, the investigator (or his designee) will call the IxRS to obtain the screening number for the patient prior to Cycle 1, Day 1.

Results of standard of care tests or examinations performed prior to obtaining informed consent and within 28 days prior to study start may be used; such tests do not need to be repeated for screening.

All screening evaluations must be completed and reviewed to confirm that patients meet all eligibility criteria before study start. The investigator will maintain a screening log to record details of all patients screened and to confirm eligibility or record reasons for screening failure, as applicable.

Patients who are on the MTD dose established in Cohort 1 must re-consent to be enrolled into Phase II.

The IxRS will be available 24 hours a day, 7 days a week. Detailed instructions regarding the IxRS will be provided to each study center. The screening numbers are to be allocated according to the specification document agreed with the IxRS provider.

Please see Appendix 1 for the schedule of screening assessments.

## 4.4.2.2 Assessments During Treatment

## For mBC Patients

Scheduled study visits are based on a q3w cycle, with Cycle 1 beginning at Day 1. All visits must occur within ± 3 business days from the scheduled date, unless otherwise noted in the schedule of assessments. All assessments will be performed on the day of the specified visit unless a time window is specified. Assessments scheduled on the day of study treatment administration should be performed prior to study treatment administration unless otherwise noted. If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend, it should be performed on the nearest following date (i.e. within 3 business days).

Local laboratory assessments scheduled for Day 1 of all cycles must be performed within 72 hours prior to study treatment administration unless

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 1

otherwise specified. Results of local laboratory assessments must be reviewed and the review documented prior to study treatment administration.

Please see Appendix 1 for the schedule of treatment period assessments.

# For mGC patients:

Scheduled study visits are based on a qw cycle, with Cycle 1 beginning at Day 1. All visits must occur within ± 3 business days from the scheduled date, unless otherwise noted in the schedule of assessments. All assessments will be performed on the day of the specified visit unless a time window is specified. Assessments scheduled on the day of study treatment administration should be performed prior to study treatment administration unless otherwise noted. If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend, it should be performed on the nearest following date (i.e. within 3 business days).

Local laboratory assessments scheduled for Day 1 of all cycles must be performed within 72 hours prior to study treatment administration unless otherwise specified. Results of local laboratory assessments must be reviewed and the review documented prior to study treatment administration.

Please see Appendix 1 for the schedule of treatment period assessments.

# 4.4.2.3 Assessments at Study Completion/Early Termination Visit

Patients may remain on study treatment until disease progression as assessed by the investigator, intolerable toxicity or the patient wishes to withdraw from study treatment. Patients who discontinue study treatment will be asked to return to the clinic approximately 28–42 days after the last study treatment administration, for the safety follow-up visit.

Please see Appendix 1 for assessments to be performed at the safety followup visit.

# 4.4.2.4 Follow-Up Assessments

After the Study Treatment Discontinuation Visit, all patients (regardless of reason for discontinuation) will have anti-cancer therapies recorded and will be followed for all unresolved study-related AEs and serious adverse events (SAEs) until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.

Patients who discontinue study drugs for any reason other than disease progression or withdrawal of consent (e.g., an AE) will continue to be followed until the development of disease progression, consent withdrawal, lost to follow-up or beginning of another anti-cancer therapy.

After the study completion/early termination visit, AEs should be followed as outlined in Section 5.5 and 5.6.

Please see Appendix 1 for the schedule of follow-up assessments.

# 4.4.2.5 Assessments at Unplanned Visits

In case unplanned visits are required, electronic Case Report Form (eCRF) pages will be available to report the information collected during those visits.

# 4.5 PATIENT, STUDY, AND SITE DISCONTINUATION

## 4.5.1 PATIENT DISCONTINUATION

Patients have the right to withdraw from the study at any time for any reason. The investigator has the right to discontinue a patient from study treatment or from the study for any medical condition that the investigator determines may jeopardize the patient's safety if he or she continues in the study, for reasons of noncompliance (e.g., missed doses, visits), if the patient becomes pregnant, or if the investigator determines it is in the best interest of the patient.

Patients must be withdrawn from study treatment if they experience any of the following:

- Pregnancy
- Disease progression defined using RECIST v. 1.1 Appendix 3. The exception to this is patients who develop isolated progression in the brain as described in Appendix 3
- Unacceptable toxicity because of the trastuzumab emtansine dose as specified in Section 5.1
- Unacceptable toxicity because of the capecitabine dose as specified in Section 5.1

Other reasons for patient discontinuation may include, but are not limited to, the following:

- Noncompliance
- Investigator decision based on the patient's best interest
- Patient decision

Patients who discontinue from study treatment prematurely for any of the above reasons will continue to be followed according to Section 4.4.2.4 "Follow-Up assessments". The primary reason for discontinuation must be recorded on the appropriate eCRF page.

## 4.5.2 STUDY DISCONTINUATION

Section 3.1.1 describes the end of study definition and discontinuation of study. Prior to that, the Sponsor has the right to terminate this study at any time. Reasons for terminating the study may include, but are not limited to, the following:

- The incidence or severity of AEs in this or other studies indicates a potential health hazard to patients
- Patient enrollment is unsatisfactory

Data recording is inaccurate or incomplete

# 5. ASSESSMENT OF SAFETY

Overall safety will be assessed on an ongoing basis during the conduct of the study.

# 5.1 SAFETY PLAN

The safety plan for patients receiving trastuzumab emtansine is based on the toxicities of trastuzumab emtansine observed in nonclinical studies; the toxicities related to its components (trastuzumab and maytansine, the parent drug of DM1) observed in clinical studies; and the clinical experience with this molecule in completed and ongoing studies. Please refer to the trastuzumab emtansine and capecitabine (Xeloda®) Investigator's Brochures for the most recent information.

All patients will be monitored closely for toxicity. The potential safety issues anticipated in this trial, as well as measures intended to avoid or minimize such toxicities, are outlined in the following sections.

#### 5.1.1 RISKS ASSOCIATED WITH TRASTUZUMAB EMTANSINE

Trastuzumab emtansine dose modifications are described in Section 5.1.5.1.

The following summarizes the experience with trastuzumab emtansine in multiple breast cancer studies to date. Trastuzumab emtansine has demonstrated a favorable toxicity and tolerability profile to date across multiple studies. Please refer to the Investigator's Brochure for further information.

Reversible thrombocytopenia has been commonly observed in completed and ongoing studies with trastuzumab emtansine. Most events were Grade 1–2; Grade 3–4 thrombocytopenia has been observed less commonly. The incidence of Grade 1 thrombocytopenia gradually increased over successive cycles; however, there was no increase in the proportion of Grade  $\geq$  3 abnormalities. The number of patients who experienced platelet count recovery to normal levels by Day 1 of the subsequent cycle decreased with successive cycles, suggesting a modest cumulative effect of trastuzumab emtansine on platelet count. There was no clear association between thrombocytopenia and severe hemorrhagic events; however, the use of platelet transfusions has been reported.

Transient and reversible increases in serum AST and ALT have been observed across the trastuzumab emtansine studies. Grade 1–2 events have been observed frequently; Grade 3–4 events have been observed much less commonly. The incidence of increased AST was substantially higher than that for ALT. Increases in AST and ALT were commonly observed by Day 8 of each cycle and generally returned to baseline by Day 21. The proportion of patients with Grade 1–2 increases in transaminases increased with successive cycles; however, no increase in the proportion of Grade 3 abnormalities over time was observed. To date, there have been no cases

meeting Hy's Law criteria for drug-induced liver injury. Although significant hepatotoxicity has rarely been seen in clinical trials with trastuzumab emtansine to date, the relationship to trastuzumab emtansine has not been established. Nevertheless, severe liver injury remains an important potential risk.

Infusion-related reactions are known to occur with the administration of monoclonal antibodies and have been reported with trastuzumab emtansine. Infusion reaction AEs occurred rarely and were mostly Grade 1–2. Non-specific symptoms that occurred on the first day of trastuzumab emtansine infusion that could be associated with an infusion reaction included fatigue, nausea, chills, pyrexia, and, less commonly, headache, hypertension, vomiting, and cough.

Pneumonitis has been rarely reported with trastuzumab emtansine. Signs, symptoms, and clinical findings include dyspnea, cough, fatigue, and pulmonary infiltrates. There were no fatalities among the cases of pneumonitis reported with trastuzumab emtansine.

In clinical trials with trastuzumab emtansine, peripheral neuropathy has been reported, mainly as Grade 1 toxicity. Hypokalemia and decreases in serum potassium have been reported in completed and ongoing studies with trastuzumab emtansine. Most of these AEs were Grade 1–2.

Although significant cardiac events have been infrequent in clinical trials with trastuzumab emtansine to date, severe cardiotoxicity remains an important potential risk. Treatment with trastuzumab, a component of trastuzumab emtansine, has resulted in subclinical and clinical cardiac failure manifesting as CHF, decreased LVEF, and cardiac death. The incidence and severity of cardiac dysfunction was highest in patients who received trastuzumab concurrently with anthracycline-containing chemotherapy regimens. Cardiotoxicity, manifesting as a decline in LVEF or CHF, is being closely monitored in the trastuzumab development program. Across studies TDM4258g, TDM4374g, and TDM4688g, approximately 273 patients were treated, and a total of 8 patients recorded an asymptomatic decrease in baseline LVEF of at least 10%, concomitant with an LVEF < 50%. Two patients had trastuzumab emtasine treatment withdrawn because of decreased LVEF. Rare cases of Grade 3 cardiac dysrhythmias have been reported among patients receiving trastuzumab emtansine, although a direct relationship to study drug remains unclear.

Importantly, preliminary evaluations of safety in the randomized study TDM4450g suggest that the safety and tolerability of trastuzumab emtansine compared favorably with that of trastuzumab plus docetaxel, with the overall incidence of Grade ≥ 3 AEs favoring the trastuzumab emtansine arm (46.4% vs. 89.4%) (data on file).

Full details regarding the clinical safety of trastuzumab emtansine are presented in Sections 5 and 6 of the Investigator's Brochure.

# 5.1.2 RISKS ASSOCIATED WITH CAPECITABINE

Capecitabine dose modifications will be done according to Section 3.1.1, study design.

Patients treated with capecitabine should be carefully monitored for toxicity. Most AEs are reversible and do not require permanent discontinuation of therapy (please refer to the Xeloda<sup>®</sup> Investigator`s Brochure for more information).

The spectrum of cardiotoxicity observed with capecitabine is similar to that of other fluorinated pyrimidines. This includes myocardial infarction, angina, dysrhythmias, cardiac arrest, cardiac failure and electrocardiographic changes. These AEs may be more common in patients with a prior history of coronary artery disease.

DPD deficiency, a rarely, unexpected, severe toxicity (e.g. stomatitis, diarrhea, neutropenia and neurotoxicity) associated with 5-FU has been attributed to a deficiency of dihydropyrimidine dehydrogenase (DPD) activity. Therefore, a link between decreased levels of DPD and increased, potentially fatal toxic effects of 5-FU cannot be excluded.

Capecitabine can induce hand–foot syndrome (palmar-plantar erythrodysesthesia or chemotherapy-induced acral erythema), which is a cutaneous toxicity. For patients receiving capecitabine monotherapy in the metastatic setting, the median time to onset was 79 days (range 11 to 360 days), with a severity range of Grades 1 to 3. Grade 1 hand-foot syndrome is defined by numbness, dysesthesia/paresthesia, tingling or erythema of the hands and/or feet and/or discomfort which does not disrupt normal activities. Grade 2 is defined as painful erythema and swelling of the hands and/or feet and/or discomfort affecting the patient's activities of daily living (ADL). Grade 3 is defined as moist desquamation, ulceration, blistering or severe pain of the hands and/or feet and/or severe discomfort that causes the patient to be unable to work or perform ADL. If Grade 2 or 3 hand-foot syndrome occurs, administration of capecitabine should be interrupted until the event resolves or decreases in intensity to Grade 1. Following Grade 3 hand-foot syndrome, subsequent doses of capecitabine should be decreased.

Capecitabine can induce hyperbilirubinemia. Administration of capecitabine should be interrupted if treatment-related elevations in bilirubin of >  $3.0 \times ULN$  or treatment-related elevations in hepatic aminotransferases (ALT, AST) of >  $2.5 \times ULN$  occur. Treatment may be resumed when bilirubin decreases to  $\leq 3.0 \times ULN$  or hepatic aminotransferases decrease to  $\leq 2.5 \times ULN$ .

# 5.1.3 TRASTUZUMAB EMTANSINE AND CAPECITABINE COMBINATION:

DLTs for the combination of trastuzumab emtansine and capecitabine will be observed during Cycle 1 (Day 1–21) of this study.

## 5.1.4 DEFINITION OF DOSE LIMITING TOXICITY

DLT toxicities will be observed during Cycle 1 (Day 1–21).
#### **Definition of DLT:**

#### Hematologic

- Uncomplicated thrombocytopenia Grade 4 which does not recover to ≥ 75.000/MI before Day 21
- 2. Thrombocytopenia (any grade) complicated with clinically significant bleeding requiring medical intervention such as: platelet transfusion, cauterization, patients with epistaxis Grade 1 or 2 may have cauterization and this should not be consider as DLT etc.
- 3. Neutropenia Grade 4 lasting > 7 consecutive days
- 4. Febrile neutropenia with an ANC of < 1000

#### Non-hematologic

- 5. Diarrhea Grade ≥ 3 which does not decrease to ≤ Grade 2 after 24 hours of starting recommended anti-diarrheal treatment in absence of DPD deficiency
- 6. Hand-foot syndrome Grade ≥ 3 in absence of DPD deficiency
- 7. Any other treatment-related toxicity ≥ Grade 3 prohibiting the start of the 2nd cycle on day 22 (3 weeks cycle length plus 1 day)
- 8. Grade 2 toxicity requiring interruption of treatment for > 7 days

NOTE: Patients experiencing ≥ Grade 3 hand-foot syndrome or diarrhea or mucositis or Febrile neutropenia with ANC < 500 during Cycle 1 must be tested for DPD deficiency (central lab will be appointed).

NOTE TO point 7, if a Grade 2 event requires a dose delay, it will not be considered as DLT.

#### 5.1.5 MANAGEMENT OF SPECIFIC ADVERSE EVENTS

#### 5.1.5.1 Trastuzumab Emtansine Dosage Modification

Patients should be assessed for toxicity prior to each dose; dosing will occur only if the clinical assessment and laboratory test values are acceptable.

Dose delays and reductions are designed to maximize treatment for those who derive clinical benefit from treatment while ensuring patient safety.

Dose delays for trastuzumab emtansine related toxicity other than the ones specified below (i.e., infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, and cardiotoxicity) are as follows:

• If significant trastuzumab emtansine related toxicities (other than infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, and cardiotoxicity) have not recovered to Grade 1 or baseline, the next scheduled dose may be delayed for up to 42 days from the last dose received. "Significant" and "related" will be based on the judgment of the investigator (in consultation with the Sponsor's Medical Monitor or designee when appropriate). For example, alopecia even if considered

- related would most likely not be considered to be significant. Fatigue may or may not be considered either related or significant.
- In general, when the significant and related toxicity (or any other toxicity that the investigator chooses to delay dosing for) resolves to Grade 1 or baseline, the patient may resume trastuzumab emtansine if the delay has not exceeded 42 days from the last received dose. Patients should be reevaluated qw during the delay, whenever possible. If dosing resumes, the patient may receive trastuzumab emtansine either at the same dose level as before or at one dose level lower than the previous dose (see Table 2 and Table 3), at the discretion of the investigator. Subsequent cycles should remain the same (q3w or qw), and patients should be assessed for toxicity.
- If a patient requires a dose reduction, dosing will be reduced by one dose level, per Table 2 or Table 3. No dose re-escalation will be allowed.
- If toxicity does not resolve within 42 days from the last dose received, the
  patient will be discontinued from study treatment and will be followed for
  disease progression and survival.
- Patients who experience a Grade 3 or 4 hematologic event should be checked at least qw for recovery. If values do not recover to baseline or Grade ≤ 1 within 42 days from the last dose received, the patient will be discontinued from study treatment.

 Table 2
 Dose Reductions for Trastuzumab Emtansine (mBC Patients)

| Dose Level | q3w Schedule |
|---------------------------------------|---------------------|
| 0 | 3.6 mg/kg |
| - 1 | 3.0 mg/kg |
| - 2 | 2.4 mg/kg |
| Indication for further dose reduction | Off study treatment |

q3w = every 3 weeks

Table 3 Dose Reductions for Trastuzumab Emtansine (mGC Patients)

| Dose Level | qw Schedule |
|---------------------------------------|-------------|
| 0 | 2.4 mg/kg |
| - 1 | 2 mg/kg |
| - 2 | Off study |
| Indication for further dose reduction | Off study |

qw = weekly

Protocol requirements for specific toxicities are outlined below.

#### Trastuzumab Emtansine Dose Modification for Thrombocytopenia

Patients receiving trastuzumab emtansine who experience any of the following events listed below, after adequate recovery to a platelet count of

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 1

Grade  $\leq$  1 (  $\geq$  75,000/µL), may continue treatment with trastuzumab emtansine at one dose level reduction in subsequent treatment cycles (see Table 2 and Table 3).

#### Grade 4 Thrombocytopenia:

Hold study drug until platelet count qualifies for Grade ≤ 1 (≥ 75,000 µL).

- Platelets < 10,000 cells/mm<sup>3</sup> for any duration
- Platelets ≥ 10,000 cells/mm³ but < 25,000 cells/mm³ for more than 7 days

#### **Grade 3 Thrombocytopenia:**

Hold study drug until platelet count qualifies for Grade  $\leq 1$  (  $\geq 75,000 \mu L$ ).

- Trastuzumab emtansine 2.4 mg/mg/week dosing
  - –Platelets must be ≥ 75,000  $\mu$ L on day of treatment.
- Trastuzumab emtansine 3.6 mg/kg/q3w dosing:
  - –Platelets must be ≥ 75,000  $\mu$ L on day of treatment.

#### **Patients on Anticoagulation Therapy:**

Hold study drug until platelet count qualifies for Grade ≤ 1 (≥ 75,000 µL).

For platelet count of Grade ≥ 3 (< 50,000 cells/µL) of any duration</li>
 Patients who experience any of these toxicities should be reassessed at least qw for recovery.

#### Trastuzumab Emtansine Dose Modification for Hepatotoxicity

Table 4 and Table 5 describe the dose modification guidelines for increases in serum bilirubin and transaminases, respectively. Patients who develop a Grade 4 serum total bilirubin increase or a Grade 4 ALT and/or AST increase must discontinue study treatment permanently. Patients should be checked assessed at least qw for the recovery of total bilirubin and/or ALT and/or AST. If total bilirubin and/or ALT and/or AST do not recover to baseline or Grade ≤ 1 (total bilirubin) or Grade ≤ 2 (ALT and/or AST) within 42 days after the last dose received, the patient must discontinue study treatment. Please see Section 5.2.3 and Table 4 and Table 5 for further information.

No re-escalation of the trastuzumab emtansine dose is allowed.

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| | Up to<br>1.5 × ULN | > 1.5–3 × ULN | ≥ 3–10 × ULN | ≥ 10 × ULN |
| T-DM1<br>action | Treat without<br>dose reduction<br>or delay | Hold <sup>a</sup> dose; reduce one dose level when recovered to Grade ≤ 1. Discontinue <sup>b</sup> if > 2 × ULN and occurs concurrent <sup>c</sup> with ALT and/or AST elevation > 3 × ULN | Hold <sup>a</sup> dose; reduce<br>one dose level when<br>recovered to<br>Grade ≤ 1.<br>Discontinue <sup>b</sup> if occurs<br>concurrent <sup>c</sup> with ALT<br>and/or AST elevation<br>> 3 × ULN | Discontinue. |

T-DM1 = trastuzumab emtansine; ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

- <sup>a</sup> A dose delay of up to 42 days after the last received dose is permitted for patients on a q3w schedule or 28 days for patients on a weekly schedule.
- <sup>b</sup> Unless a decision is made to hold then continue trastuzumab emtansine treatment based on the results of further evaluation of the situation and agreement by the investigator and the Sponsor. See also Section 5.2.3
- <sup>c</sup> Within 21 days.

Table 5 Trastuzumab Emtansine Dose Modification: Serum ALT or AST

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| | Up to<br>3 × ULN | > 3–5 × ULN | ≥ 5–20 × ULN | ≥ 20 × ULN |
| T-<br>DM1<br>action | Treat without<br>dose<br>reduction or<br>delay | Treat without dose reduction or delay. Discontinue b if occurs concurrent with total bilirubin > 2 × ULN or clinical jaundice | Hold <sup>a</sup> dose; reduce one dose level when recovered to Grade ≤ 2. Discontinue <sup>b</sup> if occurs concurrent <sup>c</sup> with total bilirubin > 2 × ULN or clinical jaundice | Discontinue |

T-DM1 = trastuzumab emtansine; ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

- <sup>a</sup> A dose delay of up to 42 days after the last received dose is permitted for patients on a q3w schedule or 28 days for patients on a weekly schedule.
- <sup>b</sup> Unless a decision is made to hold then continue trastuzumab emtansine treatment based on the results of further evaluation of the situation and agreement by the investigator and the Sponsor. See also Section 5.2.3
- <sup>c</sup> Within 21 days.

#### **Trastuzumab Emtansine Dose Modification for Neurotoxicity**

DM1, an anti-microtubule agent, can potentially cause peripheral neuropathy. Patients should be examined for signs of peripheral neuropathy prior to each dose of trastuzumab emtansine. Patients who experience Grade  $\geq 3$  neurotoxicity in the form of peripheral neuropathy that does not resolve to Grade  $\leq 2$  within 42 days after last dose received will be discontinued from study treatment.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 1

Patients receiving trastuzumab emtansine who experience Grade 3 or 4 peripheral neuropathy that does not resolve to Grade ≤ 2 within 42 days after the last dose received will be discontinued from study treatment.

#### Trastuzumab Emtansine Dose Modification for Cardiotoxicity

Patients without significant cardiac history and with a baseline LVEF ≥ 50% as determined by ECHO or MUGA scan are eligible for study participation. Ejection fractions will be monitored according to the schedules of assessment in Appendix 1.

Figure 6 summarizes the management of trastuzumab emtansine on the basis of measured LVEF and changes in LVEF from baseline. If the LVEF is reported as a range, the median of the range should be taken. If an investigator is concerned that an AE may be related to cardiac dysfunction, an additional LVEF measurement may be performed. Trastuzumab emtansine will be discontinued in any patient who develops symptomatic CHF. CHF should be treated and monitored according to standard medical practice.

The decision to stop or continue trastuzumab emtansine should be based on the algorithm shown in Figure 6. Trastuzumab emtansine must be discontinued in all patients for whom a confirmed drop of LVEF to below 40% is documented (with a repeat assessment within 21 days). For patients whose LVEF drops to values between 40% and 45% with an absolute decrease in LVEF of ≥ 10% points from baseline, trastuzumab emtansine should be held. For these patients, the LVEF should be repeated in 21 days, and trastuzumab emtansine should be discontinued if the LVEF has not recovered to within 10% absolute difference below baseline. If clinically significant cardiac dysfunction or cardiac failure develops or persists or if significant medical management is required to maintain ejection fraction, the patient should be discontinued from study treatment.

Figure 6 Algorithm for Continuation and Discontinuation of Trastuzumab Emtansine Based on Left Ventricular Ejection Fraction Assessments in Patients



CHF = congestive heart failure; LVEF = left ventricular ejection fraction.

Note: LVEF assessment results must be reviewed before the next scheduled trastuzumab emtansine infusion.

- <sup>a</sup> LVEF can be repeated within 21 days, and trastuzumab emtansine should be discontinued if LVEF < 40% is confirmed. Trastuzumab emtansine should be held while the repeat LVEF is obtained.
- After a second consecutive confirmatory result, trastuzumab emtansine should be discontinued if the LVEF is confirmed to be ≥ 10% points below baseline or if medical management was required to correct the LVEF.

## Trastuzumab Emtansine Dose Modification/Management for Infusion Reactions

No pre-medication for the first infusion of trastuzumab emtansine is required; however, pre-medication is allowed at the investigator's discretion. Patients who experience trastuzumab emtansine infusion-related temperature elevations of > 38.5°C or other minor infusion-related symptoms may be treated symptomatically with acetaminophen and/or H1 and H2 receptor antagonists (e.g., diphenhydramine and ranitidine, respectively). Serious infusion-related events (Grade ≥ 3 allergic reaction or acute respiratory distress syndrome [ARDS]) manifested by dyspnea, hypotension, wheezing, bronchospasm, tachycardia, reduced oxygen saturation, or respiratory distress should be managed with supportive therapies as clinically indicated according to standard clinical practice. Patients who experience a Grade ≥ 3 allergic reaction or ARDS will be discontinued from study treatment. Patients who have infusion-related symptoms, such as chills or fever, may have the infusion rate decreased by 50% or interrupted. When symptoms have resolved, the infusion may be restarted at ≤ 50% of the prior rate and increased in 50% increments every 30 minutes as tolerated. Pre-medication

### **Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 1

may be used before subsequent infusions at the investigator's discretion. Patients should be monitored until complete resolution of symptoms.

#### 5.1.5.2 Capecitabine Dosage Modification

#### Phase I: mBC Patients

Capecitabine dose modifications during Phase I will be performed according to the description in Section 3.1.1, study design for mBC patients.

#### Phase II: Exploration of Efficacy: mBC

During Phase II, capecitabine will be modified as per the Xeloda<sup>®</sup> Investigator's Brochure (or SMPC).

#### Phase I: mGC Patients

Capecitabine dose modifications during Phase I will be performed according to the description in Section 3.1.1, study design for mGC patients.

#### 5.2 SAFETY PARAMETERS AND DEFINITIONS

Safety assessments will consist of monitoring and recording protocol-defined AEs and SAEs; measurement of protocol-specified hematology, clinical chemistry, and urinalysis variables; measurement of protocol-specified vital signs; and other protocol-specified tests that are deemed critical to the safety evaluation of the study drug(s).

The Sponsor or its designee is responsible for reporting relevant SAEs to the Competent Authority, other applicable regulatory authorities, and participating investigators, in accordance with International Conference on Harmonisation (ICH) guidelines, Food and Drug Administration (FDA) regulations, European Clinical Trials Directive (Directive 2001/20/EC), and/or local regulatory requirements.

The Sponsor or its designee is responsible for reporting unexpected fatal or life-threatening events associated with the use of the study drug to the regulatory agencies and competent authorities by telephone or fax within 7 calendar days after being notified of the event. The Sponsor or its designee will report other relevant SAEs associated with the use of the study medication to the appropriate competent authorities (according to local guidelines), investigators, and central Institutional Review Boards/Ethics Committees (IRBs/ECs) by a written safety report within 15 calendar days of notification.

#### 5.2.1 ADVERSE EVENTS

According to the ICH guideline for Good Clinical Practice, an AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any of the following:

- Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
- Any new disease or exacerbation of an existing disease (a worsening in the character, frequency, or severity of a known condition), except as described in Section 5.3.5.7
- Recurrence of an intermittent medical condition (e.g., headache) not present at baseline
- Any deterioration in a laboratory value or other clinical test (e.g., ECG, X ray) that is associated with symptoms or leads to a change in study treatment or concomitant treatment or discontinuation from study drug
- AEs that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment (e.g., screening invasive procedures such as biopsies)

## 5.2.2 SERIOUS ADVERSE EVENTS (IMMEDIATELY REPORTABLE TO THE SPONSOR)

A SAE is any AE that meets any of the following criteria:

- Fatal (i.e., the AE actually causes or leads to death)
- Life threatening (i.e., the AE, in the view of the investigator, places the patient at immediate risk of death)

This does not include any AE that had it occurred in a more severe form or was allowed to continue might have caused death.

- Requires or prolongs inpatient hospitalization (see Section 5.3.5.8)
- Results in persistent or significant disability/incapacity (i.e., the AE results in substantial disruption of the patient's ability to conduct normal life functions)
- Congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug
- Significant medical event in the investigator's judgment (e.g., may jeopardize the patient or may require medical/surgical intervention to prevent one of the outcomes listed above)

The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an AE (rated as mild, moderate, or severe, or according to NCI CTCAE criteria; see Section 5.3.3); the event itself may be of relatively minor medical significance (such as severe headache without any further findings).

Severity and seriousness need to be independently assessed for each AE recorded on the eCRF.

SAEs are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2 for reporting instructions).

## 5.2.3 PROTOCOL-DEFINED EVENTS OF SPECIAL INTEREST/NON-SERIOUS EXPEDITED ADVERSE EVENTS

Non-serious AEs of special interest are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2 for reporting instructions). AEs of special interest for this study include the following:

Potential Drug-induced liver injury

Any potential case of drug-induced liver injury as assessed by laboratory criteria for Hy's Law will be considered as a protocol-defined event of special interest and will need to be reported to the Sponsor expeditiously. The following laboratory abnormalities define potential Hy's Law cases:

AST or ALT elevations that are > 3 × the ULN

Concurrent elevation (within 21 days of AST and/or ALT elevations) of total bilirubin > 2 × the ULN, except in patients with documented Gilbert syndrome

#### 5.2.4 PREGNANCY AND CONTRACEPTION

ICH M3 guidance requires precautions to be taken to minimize risk to fetus or embryo when including women of childbearing potential in clinical studies. These precautions include the use of highly effective contraceptive measures, excluding pregnancy at baseline (serum test), continued pregnancy monitoring, and continued pregnancy testing for up to 6 months following last dose of study drug (follow-up period based on PK considerations).

Trastuzumab, a component of trastuzumab emtansine, can cause fetal harm when administered to a pregnant woman; postmarketing case reports indicate that its use during pregnancy increases the risk for oligohydramnios during the second and third trimester. Trastuzumab has also been associated with fetal pulmonary hypoplasia, skeletal abnormalities, and neonatal death (see the Herceptin<sup>®</sup> Package Insert). There are no clinical studies of trastuzumab in pregnant women. IgGs are known to cross the placental barrier.

Therefore, trastuzumab emtansine should be not used during pregnancy. Women of childbearing potential (who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy) and men with partners of childbearing potential must agree to use a highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the patient and/or partner.

Methods of birth control which result in a low failure rate (i.e., < 1% per year) when used consistently and correctly are considered highly effective forms of contraception. The use of the following non-hormonal methods of contraception is acceptable:

 True abstinence, when this is the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, and symptothermal post ovulation methods) and withdrawal are not acceptable methods of contraception  Male sterilization (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female patients, the vasectomized male partner should be the sole partner

Alternatively, use of two of the following effective forms of contraception is acceptable:

- Placement of intrauterine device (IUD) or intrauterine system (IUS).
   Consideration should be given to the type of device being used, as there are higher failure rates for certain types (e.g., steel or copper wire)
- Condom with spermicidal foam/gel/film/cream/suppository
- Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

The use of barrier contraceptives should always be supplemented with the use of a spermicide. The following should be noted:

- Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection
- However, spermicides alone are ineffective at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone

It should be noted that two forms of effective contraception are required. A double barrier method, defined as condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, is acceptable.

Contraception is not a requirement in the case of any of the following:

- The female patient or female partner of a male patient is considered not to be of childbearing potential: if she is postmenopausal, defined by amenorrhea of ≥ 12 months duration in a woman > 45 years old; or is ≥ 40 years of age and has had amenorrhea of ≥ 24 months duration; or has undergone surgical sterilization (hysterectomy and/or bilateral oophorectomy)
- The male patient or male partner of a female patient is surgically sterilized

For male patients with a female partner of childbearing potential, cooperation of female partner is required (i.e., use of two forms of contraception as stated above) during the study and for at least 6 months following the last dose of study treatment when a highly effective form of contraception is not appropriate.

Based on PK considerations, contraception must continue for the duration of study treatment and for at least 6 months after the last dose of study treatment.

A female patient who becomes pregnant during the study must be instructed to stop taking the study medication and immediately inform the investigator. The investigator should report all pregnancies within 24 hours to the Sponsor

including the partners of male patients. The investigator should counsel the patient/partner, and discuss the risks of continuing with the pregnancy and the possible effects on the fetus. Monitoring of the patient/partner should continue until conclusion of the pregnancy. Pregnancies occurring up to 6 months after the completion of study medication must also be reported to the investigator. Please refer to Section 5.4.3 for reporting procedures.

It is not known whether trastuzumab or trastuzumab emtansine are excreted in human milk. Maternal IgG is excreted in milk and any of these monoclonal antibodies could harm infant growth and development; therefore, women should be advised to discontinue nursing during trastuzumab emtansine therapy and not to breastfeed for at least 6 months following the last dose of either study drug.

Experimental studies have reported that IgGs are present in both the preejaculate and the seminal plasma (Moldoveanu et al. 2005). To date, there
have been no clinical studies to assess the IgG profile in the pre-ejaculate and
seminal plasma in male patients receiving trastuzumab or trastuzumab
emtansine. Therefore, as a precaution male patients with female partners of
childbearing potential are required to use highly effective form of
contraception or use two forms of contraception as outlined above. Similarly,
vaginal absorption of trastuzumab emtansine is unknown and therefore male
patients with pregnant partners are required to use condoms for the duration
of the pregnancy, and then revert to contraceptive methods as outlined above.
This is to ensure that the fetus is not exposed to the study medication through
vaginal absorption. In addition, sperm or blood donation should not occur for
at least 6 months after the last dose of study treatment.

# 5.3 METHODS AND TIMING FOR CAPTURING AND ASSESSING SAFETY PARAMETERS

The investigator is responsible for ensuring that all AEs (see Section 5.2.1 for definition) are recorded on the AE eCRF and reported to the Sponsor in accordance with instructions provided in this section and in Sections 5.4, 5.5, and 5.6.

For each AE recorded on the AE eCRF, the investigator will make an assessment of seriousness (see Section 5.2.2, for seriousness criteria), severity (see Section 5.3.3), and causality (see Section 5.3.4).

#### 5.3.1 Adverse Event Reporting Period

Investigators will seek information on AEs at each patient contact. All AEs, whether reported by the patient or noted by study personnel, will be recorded in the patient's medical record and on the AE eCRF.

After informed consent has been obtained but prior to initiation of study drug, only SAEs caused by a protocol-mandated intervention should be reported (e.g., SAEs related to invasive procedures such as biopsies, medication washout, or no treatment run-in).

After initiation of study treatment, all AEs, regardless of relationship to study drug, will be reported until 30 days after the last administration of study drug

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 1

81

or study discontinuation/termination, whichever is later. After this period, investigators should report any deaths, SAEs, or other AEs of concern that are believed to be related to prior treatment with study drug (see Section 5.6).

#### 5.3.2 ELICITING ADVERSE EVENT INFORMATION

A consistent methodology of non-directive questioning should be adopted for eliciting AE information at all patient evaluation time points. Examples of non-directive questions include the following:

"How have you felt since your last clinic visit?"

"Have you had any new or changed health problems since you were last here?"

#### 5.3.3 ASSESSMENT OF SEVERITY OF ADVERSE EVENTS

The AE grading (severity) scale found in the NCI CTCAE (v. 4.0) will be used for assessing AE severity (see Table 6).

Table 6 Adverse Event Severity Grading Scale

| | Severity | Alternate Description <sup>a</sup> |
|---|---|---|
| Grade | | |
| 1 | Mild (apply event-specific NCI CTCAE grading criteria) | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate (apply event-specific NCI CTCAE grading criteria) | Minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL <sup>b</sup> |
| 3 | Severe (apply event-specific NCI CTCAE grading criteria) | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL <sup>c</sup> |
| 4 | Very severe, life-threatening,<br>or disabling (apply event-specific<br>NCI CTCAE grading criteria) | Life-threatening consequences; urgent intervention indicated |
| 5 | Death related to AE | |

ADL = activities of daily living; AE = adverse event; CTCAE = Common Terminology Criteria for Adverse Events; NCI = National Cancer Institute.

The NCI CTCAE v4.0 can be found at:

http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm#ctc\_40

Note: Regardless of severity, some events may also meet regulatory seriousness criteria. Refer to definition of a serious AE (see Section 5.2.2).

- <sup>a</sup> Use these alternative definitions for Grade 1, 2, 3, and 4 events when the observed or reported AE is not in the NCI CTCAE listing.
- b Instrumental ADL refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
- <sup>c</sup> Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

#### 5.3.4 ASSESSMENT OF CAUSALITY OF ADVERSE EVENTS

Investigators should use their knowledge of the patient, the circumstances surrounding the event, and an evaluation of any potential alternative causes to determine whether or not an AE is considered to be related to study drugs, indicating "yes" or "no" accordingly. To ensure consistency of causality assessments, investigators should apply the general guidelines outlined in Table 7.

## Table 7 Guidance for Causal Attribution of Adverse Event/Serious Adverse Event

Is the AE/SAE suspected to be caused by the investigational product based on facts, evidence, science-based rationales, and clinical judgment?

YES There is a plausible temporal relationship between the onset of the AE and administration of the investigational product, and the AE cannot be readily explained by the patient's clinical state, intercurrent illness, or concomitant therapies; and/or the AE follows a known pattern of response to the investigational product; and/or the AE abates or resolves upon discontinuation of the investigational product or dose reduction and, if applicable, reappears upon re-challenge.

Investigators should apply facts, evidence, or rationales based on scientific principles and clinical judgment to support a causal/contributory association with an investigational product.

#### NO AEs will be considered related, unless they fulfill the criteria as specified below.

Evidence exists that the AE has an etiology other than the investigational product (e.g., pre-existing medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the AE has no plausible temporal relationship to administration of the investigational product (e.g., cancer diagnosed 2 days after first dose of study drug).

Note: The investigator's assessment of causality for individual AE reports is part of the study documentation process. Regardless of the "Yes" or "No" causality assessment for individual AE reports, the Sponsor will promptly evaluate all reported SAEs against cumulative product experience to identify and expeditiously communicate possible new safety findings to investigators and applicable regulatory authorities. <a href="Attribution of SAEs will be reviewed on an ongoing basis">Attribution of SAEs will be reviewed on an ongoing basis</a>, and may be changed as additional clinical data emerges (e.g., reversibility of AE, new clinical findings in patient with AE, effects of retreatment, AEs in other patients).

In addition to assessing causality with respect to study drugs, investigators should also assess whether other factors (e.g., disease under study, concurrent illness, concomitant medication, or study procedure) may have caused the event, using similar guidance.

The investigator's assessment of causality for individual AE reports is part of the study documentation process. Regardless of the "Yes" or "No" causality assessment for individual AE reports, the Sponsor will promptly evaluate all reported serious AEs against cumulative product experience to identify and expeditiously communicate possible new safety findings to investigators and applicable regulatory authorities.

For patients receiving combination therapy, causality will be assessed individually for each protocol-mandated therapy.

#### 5.3.5 Procedures for Recording Adverse Events

Investigators should use correct medical terminology/concepts when recording AEs on the AE eCRF. Avoid colloquialisms and abbreviations.

There is one eCRF page for recording AEs or SAEs.

Only one AE term should be recorded in the event field on the AE eCRF.

#### 5.3.5.1 Diagnosis Versus Signs and Symptoms

#### Infusion-Related Reactions

AEs that occur during or within 24 hours after study drug infusion should be captured as individual signs and symptoms rather than a diagnosis of allergic reaction or infusion reaction.

#### Other Adverse Events

For AEs other than infusion-related reactions, a diagnosis (if known) should be recorded on the AE eCRF rather than individual signs and symptoms (e.g., record only liver failure or hepatitis rather than jaundice, asterixis, and elevated transaminases). However, if a constellation of signs and/or symptoms cannot be medically characterized as a single diagnosis or syndrome at the time of reporting, each individual event should be recorded on the AE eCRF. If a diagnosis is subsequently established, all previously reported AEs based on signs and symptoms should be nullified and replaced by one AE report based on the single diagnosis, with a starting date that corresponds to the starting date of the first symptom of the eventual diagnosis.

#### 5.3.5.2 Adverse Events Occurring Secondary to other Events

In general, AEs occurring secondary to other events (e.g., cascade events or clinical sequelae) should be identified by their primary cause. For example, if severe diarrhea is known to have resulted in dehydration, it is sufficient to record only diarrhea as an AE or SAE on the eCRF.

However, medically significant AEs occurring secondary to an initiating event that are separated in time should be recorded as independent events on the eCRF. For example, if a severe gastrointestinal hemorrhage leads to renal failure, both events should be recorded separately on the eCRF.

#### 5.3.5.3 Persistent or Recurrent Adverse Events

A persistent AE is one that extends continuously, without resolution, between patient evaluation time points. Such events should only be recorded once on the AE eCRF. The initial severity of the event should be recorded, and the severity should be updated to reflect the most extreme severity any time the event worsens. If the event becomes serious, the AE eCRF should be updated to reflect this.

A recurrent AE is one that resolves between patient evaluation time points and subsequently recurs. Each recurrence of an AE should be recorded separately on the AE eCRF.

#### 5.3.5.4 Abnormal Laboratory Values

Only clinically significant laboratory abnormalities that require active management will be recorded as AEs or SAEs on the eCRF (e.g., abnormalities that require study drug dose modification, discontinuation of study treatment, more frequent follow-up assessments, further diagnostic investigation, etc.).

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

If the clinically significant laboratory abnormality is a sign of a disease or syndrome (e.g., alkaline phosphatase and bilirubin 5 × ULN of normal associated with cholecystitis), only the diagnosis (e.g., cholecystitis) needs to be recorded on the AE eCRF.

If the clinically significant laboratory abnormality is not a sign of a disease or syndrome, the abnormality itself should be recorded as an AE or SAE on the eCRF. If the laboratory abnormality can be characterized by a precise clinical term, the clinical term should be recorded as the AE or SAE. For example, an elevated serum potassium level of 7.0 mEq/L should be recorded as "hyperkalemia."

Observations of the same clinically significant laboratory abnormality from visit to visit should not be repeatedly recorded as AEs or SAEs on the eCRF, unless their severity, seriousness, or etiology changes.

#### 5.3.5.5 Deaths

Deaths that occur during the protocol-specified AE reporting period (see Section 5.3.1), that are attributed by the investigator solely to progression of mBC or mGC should be recorded only on the Study Completion/Early Discontinuation eCRF. All other on-study deaths, regardless of relationship to study drug, must be recorded on the AE eCRF and immediately reported to the Sponsor (see Section 5.4.2). An independent monitoring committee will monitor the frequency of death from all causes.

Death should be considered an outcome and not a distinct event. The event or condition that caused or contributed to the fatal outcome should be recorded as the single medical concept on the AE eCRF. Generally, only one such event should be reported. If the cause of death is unknown and cannot be ascertained at the time of reporting, "unexplained death" should be recorded on the AE eCRF. If the cause of death later becomes available (e.g., after autopsy), "unexplained death" should be replaced by the established cause of death.

During post-study survival follow-up, deaths attributed to progression of mBC or mGC should be recorded only on the Survival eCRF.

#### 5.3.5.6 Pre-Existing Medical Conditions

A pre-existing medical condition is one that is present at the start of this study. Such conditions should be recorded on the Medical and Surgical History eCRF.

A pre-existing medical condition should be recorded as an AE <u>only</u> if the frequency, severity, or character of the condition worsens during the study. When recording such events on the AE eCRF, it is important to convey the concept that the pre-existing condition has changed by including applicable descriptors (e.g., "more frequent headaches").

#### 5.3.5.7 Lack of Efficacy or Clinical Worsening

Events that are clearly consistent with the expected pattern of progression of mBC or mGC should not be recorded as AEs. These data will be captured as efficacy assessment data only. In most cases, the expected pattern of progression will be based on the RECIST criteria. In rare cases, the determination of clinical progression will be based on symptomatic deterioration. However, every effort should be made to document progression using objective criteria. If there is any uncertainty as to whether an event is due to disease progression, it should be reported as an AE.

#### 5.3.5.8 Hospitalization or Prolonged Hospitalization

Any AE that results in hospitalization or prolonged hospitalization should be documented and reported as a SAE unless specifically instructed otherwise in this protocol.

There are some hospitalization scenarios that do not require reporting as an SAE when there is no occurrence of an AE. These scenarios include a planned hospitalization or prolonged hospitalization to:

- Perform an efficacy measurement for the study
- Undergo a diagnostic or elective surgical procedure for a pre-existing medical condition that has not changed
- Receive scheduled therapy for the target disease of the study

# 5.4 IMMEDIATE REPORTING REQUIREMENTS FROM INVESTIGATOR TO THE SPONSOR

Certain events require immediate reporting to allow the Sponsor to take appropriate measures to address potential new risks in a clinical trial. The investigator must report such events to the Sponsor immediately; under no circumstances should reporting take place more than 24 hours after the investigator learns of the event. The following is a list of events that the investigator must report to the Sponsor within 24 hours after learning of the event, regardless of relationship to study drug:

- Serious adverse events (SAEs)
- Non-serious AEs of special interest
- Pregnancies

The investigator must report new significant follow-up information for these events to the Sponsor immediately (i.e., no more than 24 hours) after becoming aware of the information. New significant information includes the following:

- New signs or symptoms or a change in the diagnosis
- Significant new diagnostic test results
- Change in causality based on new information
- Change in the event's outcome, including recovery
- Additional narrative information on the clinical course of the event

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Investigators must also comply with local requirements for reporting SAEs to the local health authority and IRB/EC.

#### 5.4.1 EMERGENCY MEDICAL CONTACTS

## MEDICAL MONITOR (SPONSOR'S MEDICAL RESPONSIBLE) CONTACT INFORMATION

To ensure the safety of study patients, an Emergency Medical Call Center Help Desk will access the Sponsor Medical Emergency List, escalate emergency medical calls, provide medical translation service (if necessary), connect the investigator with a Sponsor Medical Monitor, and track all calls. The Emergency Medical Call Center Help Desk will be available 24 hours per day, 7 days per week. Toll-free numbers for the Help Desk and Medical Monitor contact information will be distributed to all investigators (see "Protocol Administrative and Contact Information and List of Investigators").

# 5.4.2 REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS AND NON-SERIOUS ADVERSE EVENTS OF SPECIAL INTEREST

For reports of SAEs and non-serious AEs of special interest, investigators should record all case details that can be gathered immediately (i.e., no more than 24 hours) on the AE eCRF and submit the report via the electronic data capture (EDC) system. A report will be generated and sent to the Sponsor Safety Risk Management by the EDC system.

In the event that the EDC system is unavailable, a paper SAE/Non-Serious AE of Special Interest CRF and Fax Coversheet should be completed and faxed to the Sponsor Safety Risk Management or its designee immediately (i.e., no more than 24 hours) after learning of the event, using the fax numbers provided to investigators (see "Protocol Administrative and Contact Information & List of Investigators"). Once the EDC system is available, all information will need to be entered and submitted via the EDC system.

#### 5.4.3 REPORTING REQUIREMENTS FOR PREGNANCIES

#### 5.4.3.1 Pregnancies in Female Patients

Female patients of childbearing potential will be instructed to immediately inform the investigator if they become pregnant during the study or within 6 months after the last dose of study drug. A Pregnancy Report eCRF should be completed by the investigator immediately (i.e., no more than 24 hours) after learning of the pregnancy and submitted via the EDC system. A Pregnancy Report will automatically be generated and sent to the Sponsor Safety Risk Management. Pregnancy should not be recorded on the AE eCRF. The investigator should have the patient discontinue the study drug and discuss with the patient the risks of the pregnancy and the possible effects on the fetus. Monitoring of the patient should continue until conclusion of the pregnancy.

In the event that the EDC system is unavailable, a Pregnancy Report worksheet and Pregnancy Fax Coversheet should be completed and faxed to the Sponsor Safety Risk Management or its designee immediately (i.e., no more than 24 hours) after learning of the pregnancy, using the fax numbers provided to investigators (see "Protocol Administrative and Contact Information & List of Investigators").

#### **5.4.3.2** Pregnancies in Female Partners of Male Patients

Male patients will be instructed through the Informed Consent Form to immediately inform the investigator if their partner becomes pregnant during the study or within 6 months after the last dose of study drug. A Pregnancy Report eCRF should be completed by the investigator immediately (i.e., no more than 24 hours) after learning of the pregnancy and submitted via the EDC system. Attempts should be made to collect and report details of the course and outcome of any pregnancy in the partner of a male patient exposed to study drug. The pregnant partner will need to sign an Authorization for Use and Disclosure of Pregnancy Health Information to allow for follow-up on her pregnancy. Once the authorization has been signed, the investigator will update the Pregnancy Report eCRF with additional information on the course and outcome of the pregnancy. An investigator who is contacted by the male patient or his pregnant partner may provide information on the risks of the pregnancy and the possible effects on the fetus, to support an informed decision in cooperation with the treating physician and/or obstetrician.

In the event that the EDC system is unavailable, follow reporting instructions provided in Section 5.4.3.1.

#### 5.4.3.3 Abortions

Any spontaneous abortion should be classified as an SAE (as the Sponsor considers spontaneous abortions to be medically significant events), recorded on the AE eCRF, and reported to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2).

#### 5.4.3.4 Congenital Anomalies/Birth Defects

Any congenital anomaly/birth defect in a child born to a female patient or female partner of a male patient exposed to study drug should be classified as an SAE, recorded on the AE eCRF, and reported to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2).

# 5.5 FOLLOW-UP OF PATIENTS AFTER ADVERSE EVENTS

#### 5.5.1 INVESTIGATOR FOLLOW-UP

The investigator should follow all unresolved AEs and until the events are resolved or stabilized, the patient is lost to follow-up, or it has been determined that the study treatment or participation is not the cause of the AE/SAE. Resolution of AEs and SAEs (with dates) should be documented on the AE

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

eCRF and in the patient's medical record to facilitate source data verification (SDV).

All pregnancies reported during the study should be followed until pregnancy outcome. If the EDC system is not available at the time of pregnancy outcome, follow reporting instructions provided in Section 5.4.3.1.

#### 5.5.2 Sponsor Follow-Up

For SAEs, non-serious AEs of special interest, and pregnancies, the Sponsor or a designee may follow-up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details and outcome information (e.g., from hospital discharge summaries, consultant reports, autopsy reports) in order to perform an independent medical assessment of the reported case.

#### 5.6 POST-STUDY ADVERSE EVENTS

At the last scheduled visit, the investigator should instruct each patient to report to the investigator any subsequent AEs that the patient's personal physician believes could be related to prior study drug treatment.

The investigator should notify the Sponsor of any death, SAE or other AE of concern occurring at any time after a patient has discontinued study participation if the event is believed to be related to prior study drug treatment or study procedures. The Sponsor should also be notified if the investigator becomes aware of the development of cancer or a congenital anomaly/birth defect in a subsequently conceived offspring of a patient that participated in this study.

The investigator should report these events to the Sponsor Safety Risk Management on the AE eCRF. If the AE eCRF is no longer available, the investigator should report the event directly to Roche/Genentech Safety Risk Management via telephone via phone at +1-888-835-2555.

# 5.7 EXPEDITED REPORTING TO HEALTH AUTHORITIES, INVESTIGATORS, INSTITUTIONAL REVIEW BOARDS, AND ETHICS COMMITTEES

To determine reporting requirements for single AE cases, the Sponsor will assess the expectedness of these events using the following reference documents:

• Trastuzumab emtansine and capecitabine Investigator's Brochures
The Sponsor will compare the severity of each event and the cumulative
event frequency reported for the study with the severity and frequency
reported in the applicable reference document.

Reporting requirements will also be based on the investigator's assessment of causality and seriousness, with allowance for upgrading by the Sponsor as needed.

The Steering Committee will closely monitor the incidence of these expected events during the study. An aggregate report of any clinically relevant

imbalances that do not favor the test product will be submitted to health authorities.

# 6. <u>STATISTICAL CONSIDERATIONS AND ANALYSIS</u> PLAN

#### Phase I: mBC Patients:

Enrollment into Cohort 1, HER2-positive mBC patients, will open first.

Enrolled patients will receive study drug until Investigator-assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician or study termination by the Sponsor.

#### Phase II: Exploration of Efficacy: mBC Patients

Phase II will include only Cohort 1, i.e. mBC patients. Patients in Cohort 1, who achieved MTD level will continue with the Phase II part to be assessed for efficacy and safety. Additional patients will be enrolled in this phase in order to achieve the required sample size for this part of the study.

Enrolled patients will receive study drug until Investigator-assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician or study termination by the Sponsor.

The final analysis of Phase II part of this study for ORR will be performed at the end of study (defined in Section 3.2).

#### Phase I: mGC Patients:

Once MTD is established for Cohort 1, enrollment of HER2-positive and locally advanced or mGC patients into Cohort 2 will be opened.

Enrolled patients will receive study drug until Investigator-assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician or study termination by the Sponsor.

#### 6.1 DETERMINATION OF SAMPLE SIZE

#### Sample Size for Phase I: mBC

This part will be based on a classical 3 by 3 Phase I design. From 3 to 18 patients might be enrolled into Cohort 1. There is no formal sample size estimation for this part.

#### Sample Size for Phase II: Exploration of Efficacy: mBC

Assuming a preferable BORR rate of 75% to 80% in Cohort 1 (mBC patients) and aiming for a precision of 8-10%, lower limit of 95% confidence interval of at least 65%, a total of 100 patients would need to be evaluable for Cohort 1.

Table 8 Sample Size Estimation for Phase II

| Total number of patients is 100 (Phase II) | |
|---|---|
| Number of Patients/<br>Response | 95% Clopper-Pearson Confidence Intervals |
| 75 patients (75%) | 65–83% |
| 80 patients (80%) | 71–87% |
| Total number of patients adjusted for 10% withdrawal rate is 110 patients | |

For example, the observed BOR of 75% could be estimated to be within 65% and 83% with a probability of 95% (Clopper-Pearson exact confidence intervals). Adjusting for a withdrawal rate of approximately 10%, 110 patients will be enrolled in this phase. Patients from the Phase I (Cohort 1), who received the same dose of study medication during Phase I as chosen dose during Phase II, will contribute to the sample size of 110 patients.

The BOR rate of 75% was chosen based on previously published data for trastuzumab and capecitabine (Tjulandin et al. 2011).

The estimation of sample size was performed by Nquery and SAS programs.

#### Sample Size for Phase I: mGC

This part will be based on a classical 3 by 3 Phase I design. From 3 to 18 patients might be enrolled into Cohort 2. There is no formal sample size estimation for this part.

#### 6.2 SUMMARIES OF CONDUCT OF STUDY

#### Phase I: mBC Patients

Due to a small sample size, per-protocol (PP) population will not be defined for the Phase I Cohort 1, however major protocol violations will be summarized for this phase. A median follow-up will be estimated for Phase I, Cohort 1.

#### Phase II: Exploration of Efficacy: mBC Patients

For Phase II, Cohort 1, the PP population will be defined (Section 6.4). A median follow-up will be estimated for Phase II, Cohort 1.

#### Phase I: mGC Patients

Due to a small sample size, PP population will not be defined for the Phase I Cohort 2, however major protocol violations will be summarized for this phase. A median follow-up will be estimated for Phase I, Cohort 2.

## 6.3 SUMMARIES OF TREATMENT GROUP COMPARABILITY

#### Phase I: mBC

As Phase I is the Dose Finding part of the study, there are no treatment group comparisons for this part of the study.

Demographics, medical history and baseline characteristics will be summarized. Continuous variable will be summarized by means of median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range while categorical variables by the number and percentage of patients in each category.

#### Phase II: mBC

Phase II includes only Cohort 1, hence treatment comparability is also not applicable for this part.

Demographics, medical history and baseline characteristics will be summarized. Continuous variable will be summarized by means of median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range while categorical variables by the number and percentage of patients in each category.

#### Phase I: mGC

As Phase I is the Dose Finding part of the study, there are no treatment group comparisons for this part of the study.

Demographics, medical history and baseline characteristics will be summarized. Continuous variable will be summarized by means of median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range while categorical variables by the number and percentage of patients in each category.

#### 6.4 EFFICACY ANALYSES

#### Phase I: mBC

The main analysis population will be the safety population including all patients who received at least one dose of study medication (trastuzumab emtansine and capecitabine).

#### Phase II: Exploration of Efficacy: mBC

The main analysis population for the efficacy analysis will be the intent-to-treat population (ITT) including all new patients enrolled in Phase II and patients from Cohort 1 who achieved the MTD level. The PP population will include all ITT patients who have at least one post-baseline tumor assessment during the Phase II and no major protocol violations which will be defined in the statistical analysis plan.

#### Phase I: mGC

The main analysis population will be the safety population including all patients who received at least one dose of study medication (trastuzumab emtansine and capecitabine).

#### 6.4.1 PRIMARY EFFICACY ENDPOINT

#### Phase I: mBC Patients

The primary objectives are reaching the MTD and establishing a safety profile.

ORR, as a main efficacy endpoint, will be assessed via BORR. The BOR is defined as the best response recorded from the date when the MTD is achieved until disease progression/recurrence (or death). The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

#### Phase II: Exploration of Efficacy: mBC Patients

The primary efficacy endpoint for Phase II is the BOR as assessed by investigators. The BOR is defined as the best response recorded from the start of this Phase II until disease progression/recurrence (or death) or for patients who were involved in Phase I of the study: the best response from the date of the MTD reached until disease progression/recurrence or death. To be assigned a status of PR or CR, i.e. to be a responder, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 28 days after the criteria for response are first met, i.e. patients need to have two consecutive assessments of PR or CR. This status will be assessed only for patients with measurable disease at baseline. Patients with non-measurable disease at baseline will be assessed for the time-to-event endpoints (e.g. PFS, OS, etc).

The number and proportions of responders and non-responders together with two-sided, 95% Clopper-Pearson confidence intervals will be presented.

#### Phase I: mGC Patients

The primary objectives are reaching the MTD and establishing a safety profile.

ORR, as a main efficacy endpoint, will be assessed via BORR. The BOR is defined as the best response recorded from the date when the MTD is achieved until disease progression/recurrence (or death). The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

#### 6.4.2 SECONDARY EFFICACY ENDPOINTS

#### Phase I: mBC

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### Phase II: Exploration of Efficacy: mBC

The secondary endpoints for Phase II will be:

- Time to response (TTR)
- Duration of response (DoR)
- Time to progression (TTP)
- Time to treatment failure (TTF)
- Progression free survival (PFS)
- Clinical benefit rate (CBR)
- Overall survival (OS)

TTR is defined as the time from enrollment to first documentation of confirmed PR or CR (whichever occurs first). Patients who do not have a confirmed response will be censored at the date of the last tumor assessment.

DoR is defined as the period from the date of initial confirmed PR or CR until the date of PD or death from any cause. Patients with no documented progression after CR or PR will be censored at the last date at which they are known to have had the CR or PR, respectively. The method for handling censoring is the same as described for the PFS below. Only patients with BOR of CR or PR (i.e. responders) will be included in the analysis of DoR.

For patients with a BOR of CR or PR, TTR is defined as the time from the date of enrollment into Cohort 1 to the date of first CR or PR. The censoring rules will be similar to those of the PFS.

TTP is defined as time from enrollment into Cohort 1 to the first occurrence of PD. Patients who have not progressed at the time of study completion (including patients who have died before PD) or who are lost to follow-up are censored at the date of the last tumor assessment.

TTF is defined from enrollment into Cohort 1 until TTF, for example, to disease progression, death, withdrawal due to AE or lab abnormality, or refusal of treatment. Patients who do not experience any of the above events while on study will be censored on the day of their last tumor assessment. For patients who were already in Phase I, the start date will be date of first study medication that was chosen for Phase II.

PFS is defined as the time from enrolment into Cohort 1 until the first documented progression of disease or death from any cause, whichever occurs first. For patients who were already enrolled in Cohort 1 during Phase 1, the time to PFS will be defined from the start date of study medication that was chosen for Phase II. Patients with no PFS events will be censored at the time of the last evaluable tumor assessment. Patients with no tumor assessment after the baseline visit at the time of Phase II will be censored at the time of enrolment plus 1 day.

Clinical benefit response includes patients whose best (confirmed) response was PR or CR or stable disease that lasts at least 6 months.

OS is defined as the time from the date of enrollment into Cohort 1 until the date of death, regardless of the cause of death. For patients who were already in Phase I, same rule as for PFS will be applied. Patients who were alive at the time of the analysis will be censored at the date of the last follow-up assessment.

Estimates for the survivor function for the time-to-event variable such as TTR, DoR, TTP, TTF, PFS, and OS, will be obtained by using the Kaplan-Meier approach. CBR will be summarized in a similar way to the primary efficacy endpoint, BOR.

#### Phase I: mGC

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### 6.5 SAFETY ANALYSES

#### Safety Population Phase I: mBC

The safety population (SP) Phase I, mBC will include all patients who received at least one dose of study medication during Phase I. Safety endpoints will be summarized for this part of the study and presented.

Safety parameters will be analysed in a similar way to safety parameters in Phase I: mGC.

#### Phase II: Exploration of Efficacy: mBC

The SP Phase II, mBC will include all patients who received at least one dose of study medication during Phase II. Safety endpoints will be summarized for this part of the study and presented.

Safety endpoints during Phase II will be assessed via: total AEs, AEs Grade ≥ 3, SAEs, premature withdrawal from study and study medication, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by MedDRA preferred term. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry, will be presented in shift tables of NCI-CTC grade at baseline *versus* worst grade during treatment for Cohort 1, Phase II and overall.

LVEF will be summarized over time by means of mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### Safety Population Phase I: mGC

The SP Phase I, mGC will include all patients who received at least one dose of study medication during Phase I. Safety endpoints will be summarized for this part of the study and presented.

Safety parameters for this part of the study will be summarized by treatment dose. The summaries of AEs, SAEs, AEs that cause discontinuation from the study treatment will be analyzed in a similar way to AEs in Phase II.

The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by MedDRA preferred term. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry, will be presented in shift tables of NCI-CTC grade at baseline *versus* worst grade during treatment for Cohort 2, Phase I and overall.

LVEF will be summarized over time by means of mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### 6.6 PHARMACODYNAMIC ANALYSES

No pharmacodynamic analyses are planned for this study.

#### 6.7 PHARMACOKINETIC ANALYSES

#### For Phase I only (mBC and mGC Patients):

The following PK parameters of trastuzumab emtansine and capecitabine (not limited to these listed) will be determined only in the Phase I part of the study for Cohort 1 and Cohort 2 in all patients who receive study treatment using either non-compartmental and/or population methods, if data allow:

- Serum concentrations of trastuzumab emtansine (conjugate) and total trastuzumab
- Plasma concentrations of DM1, capecitabine and its active metabolite 5fluorouracil (5-FU)
- Total exposure (AUC)
- C<sub>max</sub>

- Clearance (CL)
- Volume of distribution (V<sub>d</sub>)
- Terminal half-life (T<sub>1/2</sub>)

The pharmacokinetics of trastuzumab emtansine, total trastuzumab and DM1 will be compared with historical single agent PK data to evaluate the potential effect of capecitabine on the PK of trastuzumab emtansine and related analytes. The PK of capecitabine and its active metabolite 5-FU in cycle 1 (in the absence of trastuzumab emtansine) will be compared with the PK of cycle 2 (in the presence of trastuzumab emtansine) to evaluate the potential effect of trastuzumab emtansine on the PK of capecitabine and 5-FU.

All PK parameters will be listed and tabulated by treatment dose and by Cohort. Descriptive summary statistics including arithmetic mean, geometric mean (e.g. AUC and  $C_{max}$ ), median, range, SD and coefficient of variation will be presented for each cohort. Nonlinear mixed effects modeling will be also used but details will be presented in the statistical analysis plan.

#### 6.8 EXPLORATORY ANALYSES

#### For Phase II: Exploration of Efficacy in mBC Patients only:

Subgroup analysis for BOR, safety (AEs, SAEs and AE with Grade ≥ 3) in Phase II will be presented for: elderly *versus* younger patients, and patients with ECOG 0–1 *versus* ECOG 2. More details about subgroups will be provideded in the statistical analysis plan.

#### **Pharmacoeconomic Endpoint:**

The resource expenditure due to hospitalizations that are not study-defined evaluations while on study treatment will be evaluated. The number of hospital visits, number of days admitted, and type of visits (emergency department *versus* inpatient care) will be collected. The reason for admission (disease progression *versus* AE) will also be assessed.

#### 6.9 INTERIM ANALYSES

There is no formal efficacy interim analysis.

The design of this study includes: Phase I, Phase II and different cohorts. Corresponding analyses as described in the protocol will be performed when all data for particular cohort and study phase are collected and cleaned.

#### 7. DATA COLLECTION AND MANAGEMENT

#### 7.1 DATA QUALITY ASSURANCE

The Sponsor will be responsible for data management of this study, including quality checking of the data. Data entered manually will be collected via EDC using eCRFs. The sites will be responsible for data entry into the EDC system. In the event of discrepant data, the Sponsor will request data clarification from the sites, which the sites will resolve electronically in the EDC system.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

The Sponsor will produce an EDC Study Specification document that describes the quality checking to be performed on the data. Central laboratory data and other electronic data will be sent directly to the Sponsor, using the Sponsor's standard procedures to handle and process the electronic transfer of these data.

eCRFs and correction documentation will be maintained in the EDC system's audit trail. System backups for data stored by the Sponsor and records retention for the study data will be consistent with the Sponsor's standard procedures.

#### 7.2 ELECTRONIC CASE REPORT FORMS

eCRFs are to be completed using a Sponsor-designated EDC system. Sites will receive training and have access to a manual for appropriate eCRF completion. eCRFs will be submitted electronically to the Sponsor and should be handled in accordance with instructions from the Sponsor.

All eCRFs should be completed by designated, trained site staff. eCRFs should be reviewed and electronically signed and dated by the investigator or a designee.

At the end of the study, the investigator will receive patient data for his or her site in a readable format on a compact disc that must be kept with the study records. Acknowledgement of receipt of the compact disc is required.

#### 7.3 SOURCE DATA DOCUMENTATION

Study monitors will perform ongoing SDV to confirm that critical protocol data (i.e., source data) entered into the eCRFs by authorized site personnel are accurate, complete, and verifiable from source documents.

Source documents (paper or electronic) are those in which patient data are recorded and documented for the first time. They include, but are not limited to, hospital records, clinical and office charts, laboratory notes, memoranda, patient-reported outcomes, evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies of transcriptions that are certified after verification as being accurate and complete, microfiche, photographic negatives, microfilm or magnetic media, X-rays, patient files, and records kept at pharmacies, laboratories, and medico-technical departments involved in a clinical trial.

Source documents that are required to verify the validity and completeness of data entered into the eCRFs must not be obliterated or destroyed.

To facilitate SDV, the investigators and institutions must provide the Sponsor with direct access to applicable source documents and reports for trial-related monitoring, Sponsor audits, and IRB/EC review. The investigational site must also allow inspection by applicable health authorities.

#### 7.4 USE OF COMPUTERIZED SYSTEMS

When clinical observations are entered directly into an investigational site's computerized medical record system (i.e., in lieu of original hardcopy records),

**Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 1

the electronic record can serve as the source document if the system has been validated in accordance with health authority requirements pertaining to computerized systems used in clinical research. An acceptable computerized data collection system (for clinical research purposes) would be one that (1) allows data entry only by authorized individuals; (2) prevents the deletion or alteration of previously entered data and provides an audit trail for such data changes (e.g., modification of file); (3) protects the database from tampering; and (4) ensures data preservation.

In collaboration with the study monitor, Sponsor's Quality Assurance group may assist in assessing whether electronic records generated from computerized medical record systems used at investigational sites can serve as source documents for the purposes of this protocol.

If a site's computerized medical record system is not adequately validated for the purposes of clinical research (as opposed to general clinical practice), applicable hardcopy source documents must be maintained to ensure that critical protocol data entered into the eCRFs can be verified.

#### 7.5 RETENTION OF RECORDS

U.S. FDA regulations (21 Code of Federal Regulations §312.62[c]) and the ICH Guideline for Good Clinical Practice (GCP) (see Section 4.9 of the guideline) require that records and documents pertaining to the conduct of this study and the distribution of investigational drug, including eCRFs, Consent Forms, laboratory test results, and medication inventory records, must be retained by the Principal Investigator for 2 years after the last marketing application approval in an ICH region or after at least 2 years have elapsed since formal discontinuation of clinical development of the investigational product. All state and local laws for retention of records also apply.

No records should be disposed of without the written approval of the Sponsor. Written notification should be provided to the Sponsor for transfer of any records to another party or moving them to another location.

For studies conducted outside the United States under a U.S. Investigational New Drug application (IND), the Principal Investigator must comply with the record retention requirements set forth in the U.S. FDA IND regulations and the relevant national and local health authorities, whichever is longer.

#### 8. <u>ETHICAL CONSIDERATIONS</u>

#### 8.1 COMPLIANCE WITH LAWS AND REGULATIONS

This study will be conducted in full conformance with the ICH E6 guideline for GCP and the principles of the Declaration of Helsinki, or the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual. The study will comply with the requirements of the ICH E2A guideline (Clinical Safety Data Management: Definitions and Standards for Expedited Reporting). Studies conducted in the United States or under a U.S. Investigational New Drug (IND) application will comply with U.S. FDA regulations and applicable local, state, and federal laws.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Studies conducted in the European Union (EU)/European economic area (EEA) will comply with the EU Clinical Trial Directive (2001/20/EC).

#### 8.2 INFORMED CONSENT

Sponsor's sample Informed Consent Form will be provided to each site. If applicable, it will be provided in a certified translation of the local language. The Sponsor or its designee must review and approve any proposed deviations from the Sample Informed Consent Form or any alternate Consent Forms proposed by the site before IRB/EC submission. The final IRB/EC-approved Consent Forms must be provided to the Sponsor for health authority submission purposes according to local requirements.

The Consent Form must be signed and dated by the patient or the patient's legally authorized representative before his or her participation in the study. The case history or clinical records for each patient shall document the informed consent process and that written informed consent was obtained prior to participation in the study.

A copy of each signed Consent Form must be provided to the patient or the patient's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

All signed and dated Consent Forms must remain in each patient's study file and must be available for verification by study monitors at any time.

The Informed Consent Form should be revised whenever there are changes to procedures outlined in the informed consent or when new information becomes available that may affect the willingness of the patient to participate.

For any updated or revised Consent Forms, the case history for each patient shall document the informed consent process and that written informed consent was obtained for the updated/revised Consent Form for continued participation in the study. The final revised IRB/EC-approved Informed Consent Form must be provided to the Sponsor for regulatory purposes.

If the site uses a separate Authorization Form for patient authorization to use and disclose personal health information under the U.S. Health Insurance Portability and Accountability Act (HIPAA) regulations, the review, approval, and other processes outlined above apply except that IRB/IEC review and approval may not be required per study site policies.

# 8.3 INSTITUTIONAL REVIEW BOARD OR ETHICS COMMITTEE

This protocol, the Informed Consent Forms, any information to be given to the patient, and relevant supporting information must be submitted to the IRB/EC by the Principal Investigator and reviewed and approved by the IRB/EC before the study is initiated. In addition, any patient enrollment materials must be approved by the IRB/EC.

The Principal Investigator is responsible for providing written summaries of the status of the study to the IRB/EC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC. Investigators are also responsible for promptly informing the IRB/EC of any protocol amendments.

In addition to the requirements to report protocol-defined AEs to the Sponsor, investigators are required to promptly report to their respective IRB/EC all unanticipated problems involving risk to human patients. Some IRBs/ECs may want prompt notification of all SAEs, whereas others require notification only about events that are serious, assessed to be related to study treatment, and are unexpected. Investigators may receive written IND safety reports or other safety related communications from the Sponsor. Investigators are responsible for ensuring that such reports are reviewed and processed in accordance with regulatory requirements and with the policies and procedures established by their IRB/EC and archived in the site's study file.

#### 8.4 CONFIDENTIALITY

The Sponsor maintains confidentiality standards by coding each patient enrolled in the study through assignment of a unique patient identification number. This means that patient names are not included in data sets that are transmitted to any Sponsor location.

Patient medical information obtained by this study is confidential and may only be disclosed to third parties as permitted by the Informed Consent Form (or separate authorization for use and disclosure of personal health information) signed by the patient, unless permitted or required by law.

Medical information may be given to a patient's personal physician or other appropriate medical personnel responsible for the patient's welfare, for treatment purposes.

Data generated by this study must be available for inspection upon request by representatives of the U.S. FDA and other national and local health authorities, the Sponsor monitors, representatives, and collaborators, and the IRB/EC for each study site, as appropriate.

#### 8.5 FINANCIAL DISCLOSURE

Investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate health authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

# 9. <u>STUDY DOCUMENTATION, MONITORING, AND ADMINISTRATION</u>

#### 9.1 STUDY DOCUMENTATION

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented, including but not limited to the

protocol, protocol amendments, Informed Consent Forms, and documentation of IRB/EC and governmental approval. In addition, at the end of the study, the investigator will receive the patient data, which includes an audit trail containing a complete record of all changes to data.

#### 9.2 SITE INSPECTIONS

Site visits will be conducted by the Sponsor or an authorized representative for inspection of study data, patients' medical records, and eCRFs. The investigator will permit national and local health authorities, the Sponsor monitors, representatives, and collaborators, and the IRBs/ECs to inspect facilities and records relevant to this study.

#### 9.3 ADMINISTRATIVE STRUCTURE

The study will have a Steering Committee, central laboratory, IxRS, eCRF, and will be conducted by a contract research organization (CRO) together with the Sponsor.

## 9.4 PUBLICATION OF DATA AND PROTECTION OF TRADE SECRETS

The results of this study may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the Sponsor prior to submission. This allows the Sponsor to protect proprietary information and to provide comments based on information from other studies that may not yet be available to the investigator.

The Sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter trials only in their entirety and not as individual center data. In this case, a coordinating investigator will be designated by mutual agreement.

Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements. Any formal publication of the study in which contribution the Sponsor personnel exceeded that of conventional monitoring will be considered as a joint publication by the investigator and the appropriate the Sponsor personnel.

Any inventions and resulting patents, improvements, and/or know-how originating from the use of data from this study will become and remain the exclusive and unburdened property of the Sponsor, except where agreed otherwise.

#### 9.5 PROTOCOL AMENDMENTS

Any protocol amendments will be prepared by the Sponsor. Protocol amendments will be submitted to the IRB/EC and to regulatory authorities in accordance with local regulatory requirements.

Approval must be obtained from the IRB/EC and regulatory authorities (as locally required) before implementation of any changes, except for changes

necessary to eliminate an immediate hazard to patients or changes that involve logistical or administrative aspects only (e.g., change in Medical Monitor or contact information).

#### 10. REFERENCES

- 1. Albarello, L, Pecciarini, L, & Doglioni, C (2011). HER2 testing in gastric cancer. Advances in anatomic pathology 2011; 18:53–59.
- 2. Austin CD, De Mazière AM, Pisacane PI, et al. Endocytosis and sorting of ErbB2 and the site of action of cancer therapeutics trastuzumab and geldanamycin. Mol Biol Cell 2004; 15:5268-5282.
- Bang YJ, van Cutsem E, Feyereislova A, et al. Trastuzumab in combination with chemotherapy *versus* chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet 2010; 376:687–697.
- 4. Blum JL, Dieras V, Lo Russo PM, et al. Multicenter, phase II study of oral capecitabine in taxane-pretreated metastatic breast carcinoma patients. Cancer 2001; 92:1759–1768.
- 5. Blum JL, Jones SE, Buzdar AU, et al. Multicenter phase II study of capecitabine in paclitaxel-refractory metastatic breast cancer. J Clin Oncol 1999; 17:485–493.
- Cabanillas F, Chan KK, Floss HG, et al. Results of a phase II study of maytansine in patients with breast carcinoma and melanoma. Cancer Treat Rep. 1979; 63:507–9.
- 7. Cassady JM, Chan KK, Floss HG, et al. Recent developments in the maytansinoid antitumor agents. Chem Pharm Bull (Tokyo) 2004; 52:1–26.
- 8. Catalano V, Labianca R, Beretta GD, et al. Gastric cancer. Crit Rev Oncol Hematology 2005; 54:209–241.
- 9. Igawa Y, Matsubara M, Matsunaga K et al. Pharmacokinetic (PK) and pharmacodynamic (PD) analysis of trastuzumab emtansine (T-DM1) in Japanese patients with advanced or recurrent HER2-positive breast cancer (JO22591): Comparison with Western patients. ASCPT 2012.
- 10. De Vivo R, Pignata S, Palaia R, et al. The role of chemotherapy in the management of gastric cancer. J Clin Gastroenterol. 2000; 30:364–371.
- 11. Erickson HK, Park PU, Widdison WC, et al. Antibody-maytansinoid conjugates are activated in targeted cancer cells by lysosomal degradation and linker-dependent intracellular processing. Cancer Res. 2006; 66:4426–4433.
- 12. Faivre J, Forman D, Esteve J, et al. Survival of patients with oesophageal and gastric cancers in Europe. Eur J Cancer. 1998; 34:2167–2175.
- 13. Ferlay J, Shin HR, Bray F, et al. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer 2010; 127:2893–917.
- 14. Geyer CE, Forster J, Lindquist D, et al. Lapatinib plus capecitabine for HER2-positive advanced breast cancer. N Engl J Med. 2006; 355:2733–43.
- 15. Girish S, Gupta M, Wang B, et al. Clinical pharmacology of trastuzumab emtansine (T-DM1): an antibody–drug conjugate in development for the

- treatment of HER2-positive cancer. Cancer Chemother Pharmacol. 2012; 69:1229–40.
- 16. Gupta M, LoRusso PM, Wang B et al. Clinical implications of pathophysiological and demographic covariates on the population pharmacokinetics of trastuzumab-DM1, a HER2-targeted antibody–drug conjugate, in patients with HER2-positive metastatic breast cancer. J Clin Pharmacol. 2012; 52:691–703.
- 17. Hofmann M, Stoss O, Shi D, et al. Assessment of a HER2 scoring system for gastric cancer: results from a validation study. Histopathology 2008; 52:797–805.
- 18. Issell BF, Crooke ST. Maytansine. Cancer Treat Rev. 1978; 5:199–207.
- 19. Jemal A, Bray F, Center MM, et al. Global Cancer Statistics. CA Cancer J Clin. 2011; 61:69–90.
- Junttila TT, Li G, Parsons K, et al. Trastuzumab-DM1 (T-DM1) retains all the mechanisms of action of trastuzumab and efficiently inhibits growth of lapatinib insensitive breast cancer. Breast Cancer Res Treat 2011; 128:347–56.
- 21. Krop IE, Beeram M, Modi S et al. Phase I study of trastuzumab-DM1, an HER2 antibody-drug conjugate, given every three weeks to patients with HER2-positive metastatic breast cancer. J. Clin Oncol 2010; 28:2698-2704.
- 22. Krop IE, Mita M, Burris HA, et al. A Phase I Study of Weekly Dosing of Trastuzumab-DM1 (T-DM1) in Patients with Advanced HER 2-Positive Breast Cancer. Clin Oncol 2008; 26:suppl.abstract:1029.
- 23. Krop IE, Mita M, Burris HA, et al. A phase I study of weekly dosing of trastuzumab-DM1 (T-DM1) in patients with advanced HER2+ breast cancer. (SABCS 2008) Cancer Res 2009; 69:suppl1:3136.
- 24. Lewis Phillips G, Fields CT, Crocker L, et al. Potent anti-tumor activity of trastuzumab-DM1 antibody conjugate in combination with cytotoxic chemotherapeutic agents, antibodies or small molecule kinase inhibitors. AACR 2008; poster#2133.
- 25. Marty M, Cognetti F, Maraninchi D, et al. Randomized phase II trial of the efficacy and safety of trastuzumab combined with docetaxel in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer administered as first-line treatment: the M77001 study group. J Clin Oncol. 2005; 23:4265–74.
- 26. Moldoveanu Z, Huang W-Q, Kulhavy R, et al. Human male genital tract secretions: both mucosal and systemic immune compartments contribute to the humoral immunity. J Immunol 2005; 175:4127–36.
- 27. Parkin DM, Bray F, Ferlay J, et al. Global Cancer Statistics 2002. CA Cancer J Clin. 2005; 55:74–108.
- 28. Power DG, Kelsen DP, Shah MA. Power Advanced gastric cancer--slow but steady progress. Cancer Treat Rev. 2010; 36:384-92.
- 29. Press MF, Sauter G, Bernstein L, et al. Diagnostic evaluation of HER-2 as a molecular target: an assessment of accuracy and reproducibility of laboratory testing in large, prospective, randomized clinical trials. Clin Cancer Res 2005; 11:6598–607.
- Ries LAG, Melbert D, Krapcho M, et al (eds). SEER Cancer Statistics Review 1975 2005. Bethesda (MD): National Cancer Institute, 2008;http://seer.cancer.gov/csr/1975 2005
- 31. Sawaki A, Ohashi Y, Omuro Y, et al. Efficacy of trastuzumab in Japanese patients with HER2-positive advanced gastric or gastroesophageal junction cancer: a subgroup analysis of the Trastuzumab for Gastric Cancer (ToGA) study. Gastric Cancer 2011; epub ahead of print. DOI: 10.1007/s10120-011-0118-1.
- 32. Shen B-Q, Bumbaca D, Saad O, et al. Metabolic Fate and Pharmacokinetic Characterization of Trastuzumab Emtansine (T-DM1): An Emphasis on Preclinical and Clinical Catabolism. ASCPT 2011.
- 33. Slamon DJ, Clark GM, Wong SG et al. Human breast cancer; correlation of relapse and survival with amplification of the HER2/neo oncogene. Science 1987; 235:177–182.
- 34. Slamon DJ, Leyland-Jones B, Shak S, et al. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med. 2001; 344:783–92.
- 35. Spector NL, Xia W, Burris H 3<sup>rd</sup>, et al. Study of the biologic effects of lapatinib, a reversible inhibitor of ErbB1 and ErbB2 tyrosine kinases, on tumor growth and survival pathways in patients with advanced malignancies. J Clin Oncol. 2005; 23:2502–12.
- 36. Sundaresan S, Penuel E, Sliwkowski MX. The biology of human epidermal growth factor receptor 2. Curr Oncol Rep. 1999;1:16–22.
- 37. Tanner M, Hollmen M, Junttila TT, et al. Amplification of HER2 in gastric cancer—association with topoisomerase IIa gene amplification, intestinal type, poor prognosis and sensitivity to trastuzumab. Annals Oncol. 2005; 16: 273–278.
- 38. Therasse P, Eisenhauer EA, Verwij J. RECIST revisited: a review of validation studies on tumour assessment. Eur J Cancer. 2000; 42:1031–1039.
- 39. Tjulandin S, Makhson A, Gligorov J, et al. First results of a Phase II study of Bevacizumab in combination with trastuzumab and capecitabine as first-line treatment of HER2-positive LR/MBC. ASCO 2011; Poster#571.
- 40. von Minckwitz G, Schwedler K, Schmidt M, et al. Trastuzumab beyond progression: overall survival analysis of the GBG 26/BIG 3-05 phase III study in HER2-positive breast cancer. Eur J Cancer 2011; 47:2273–81.
- 41. Yang J, Wang Y, Zhao H, et al. Combination of exposure-response and case-control analyses in regulatory decision making. J Clin Oncol 2011; 29: suppl; 4087.

Trastuzumab Emtansine RO5304020

- 42. Yoon HH, Shi Q, Sukov WR, et al. Association of HER2/ErbB2 expression and gene amplification with pathologic features and prognosis in esophageal adenocarcinomas. Clin Cancer Res. 2012; 18:546-54.
- 43. Wardley A, et al. Trastuzumab plus docetaxel with or without capecitabine in patients with HER2-positive advanced/metastatic breast cancer: first efficacy results from the Phase II MO16419 (CHAT) Study. SABCS 2006; Abstract# 2063.
- 44. WHO, World Health Statistics 2011.

### Appendix 1 Schedule of Assessments

#### Table 1Schedule of assessments for mBC patients (Phase I and II, Cohort 1)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | Cycle 4 onward | | ards | Safety<br>Follow-Up<br>Visit | Safety<br>Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 6<br>months |
| Informed Consent | X <sup>a</sup> | | | | | | | | | | | |
| HER2 Status | Xp | | | | | | | | | | | |
| Medical History and Demographics | X | | | | | | | | | | | |
| Complete Physical Examination | X | | | | | | | | | | | |
| Limited Physical Examination <sup>c</sup> | | X | | | Х | | | Х | | | Х | |
| Height and Weight <sup>d</sup> | X | Х | | | Х | | | Х | | | Х | |
| Vital Signs <sup>e</sup> | X | Х | | | Х | | | Х | | | Х | |
| ECOG Performance Status | X | Х | | | Х | | | Х | | | Х | |
| Concomitant Medication Reporting | X <sup>f</sup> | Х | | | • | | Ongoii | ng | | | | |
| Adverse Event Reporting | X <sup>g</sup> | | • | | | Ongoing | | | | | Х | X <sup>h</sup> |
| 12-lead ECG | Х | | | | | | | | | | | |
| ECHO/MUGA <sup>i</sup> | X <sup>i</sup> | | | Xi | | | Xi | | | X <sup>i</sup> | X <sup>i</sup> | |
| Tumor Assessments <sup>i</sup> | Х | | At cycle 3 (9 weeks after C1 D1), and then every 4 <sup>th</sup> cycle (12 weeks there-after, regardless of dose delay or early discontinuation, until disease progression or study termination) | | | | | х | | | | |
| Brain CT or MRI <sup>k</sup> | Х | | | At the disc | retion of th | ne investig | ator, if clin | ically indic | cated, unti | l disease ¡ | progression | |
| Bone Scan/Imaging <sup>I</sup> | Х | | | | | | As clinical | y indicated | d | | | |

#### Table 1Schedule of assessments for mBC patients (Phase I and II, Cohort 1) (cont.)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | Cycl | e 4 onwa | rds | Safety<br>Follow-Up<br>Visit | Safety<br>Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 6<br>months |
| Hematology <sup>m</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | | | Х | |
| Biochemistry <sup>o</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | | | Х | |
| Urinalysis <sup>p</sup> | Х | | As clinically indicated | | | | | | Х | | | |
| INR/aPTT | Х | A | As clinically indicated, e.g. for patients receiving anticoagulation therapy | | | | | Х | | | | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Χ <sup>q</sup> | | | Χ <sup>q</sup> | Х | Х |
| PK/PD Samples (see Appendix 2) <sup>r</sup> | | X <sup>r</sup> | | | X <sup>r</sup> | | | | | | | |
| Assessment of Patient Hospitalizations and/or Hospital Visits | | Х | | | Х | | | Х | | | х | |
| Administration of trastuzumab emtansine | | D 2 <sup>s</sup> | | | D 1 <sup>s</sup> | | | D 1 <sup>s</sup> | | | | |
| Administration of capecitabine | | D 1–14 D 1–14 D 1–14 | | | | | | | | | | |
| Overall survival | Х | | X | | | | | Х | Х | | | |

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

- 1.NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within **14 days** prior to first treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1).
- 2.All patients will be followed up every 6 months (except for pregnancy every 3 months) until disease progression or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than disease progression will continue to undergo tumor assessments every 3–6 months.
- a)Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests. Patients who are on the MTD dose established in Cohort 1 must re-consent to be enrolled into Phase II.
- b)HER2-positivity is defined as IHC 3+ or gene amplification by ISH. It will be performed locally for mBC patients.
- c)Limited symptom-directed physical examination.
- d)Height to be obtained at screening or at Cycle 1 Day 1 only.
- e)Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f)Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to first study treatment.
- g)During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h)Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatment-related AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i)Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, and on Day 15-21 of Cycle 1, Cycle 3 and every third cycle thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

# Study MO28230

### Appendix 1 Schedule of Assessments (cont.)

- j)Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than disease progression, continued tumor assessments according to the protocol schedule of assessments is required.
- k)Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 4 months) as detailed in Section 4.4.1.4 of the protocol and in Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- I)An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed >28 days but ≤ 60 days prior to study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- m)Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and white blood cells (WBC) with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils.
- n)Assessments should be performed at screening, on Day 1, 8 and 15 of Cycles 1–3, on Day 1 of all subsequent cycles, and weekly following any hematologic AE. If capecitabine is discontinued due to toxicity, assessments should be performed weekly (minimum) until resolution of the AE (Grade ≤ 1/ baseline), and on Day 1 of subsequent cycles thereafter. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- o)Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, blood urea nitrogen (BUN)/urea, creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN). p)Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.

- q)Serum β-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.
- r)Pharmacokinetic assessments will be performed during the dose finding period of the study only (see Appendix 2).
- s)Trastuzumab emtansine will be administered on Day 1 of each 3 weekly cycle for all mBC patients in Cohort 1 and Phase II period of the study except in the first cycle where trastzumab emtansine will be given on DAY 2 (to allow PK sampling).

#### Table 2Schedule of assessments for mGC patients (Phase I, Cohort 2)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2-3 | 3 | Су | cle 4 onwa | ards | Safety<br>Follow-Up<br>Visit | Safety<br>Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 6<br>months |
| Informed Consent | Xª | | | | | | | | | | | |
| HER2 Status | Xp | | | | | | | | | | | |
| Medical History and Demographics | Х | | | | | | | | | | | |
| Complete Physical Examination | Х | | | | | | | | | | | |
| Limited Physical Examination <sup>c</sup> | | Х | | | Х | | | Х | | | Х | |
| Height and Weight <sup>d</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Vital Signs <sup>e</sup> | Х | Х | | | Х | | | Х | | | Х | |
| ECOG Performance Status | Х | Х | | | Х | | | Х | | | Х | |
| Concomitant Medication Reporting | X <sup>f</sup> | Х | | | | | Ongoi | ng | | | | |
| Adverse Event Reporting | X <sup>g</sup> | | | | | Ongoing | | | | | Х | X <sup>h</sup> |
| 12-lead ECG | Х | | | | | | | | | | | |
| ECHO/MUGA <sup>i</sup> | X <sup>i</sup> | | | X <sup>i</sup> | | | X <sup>i</sup> | | | Xi | X <sup>i</sup> | |
| Tumor Assessments <sup>j</sup> | Х | At 9 we | At 9 weeks after C1D1, and every 12 weeks thereafter, regardless of dose delay or early discontinuation, until disease progression or study termination | | | | | | | | | |
| Brain CT or MRI <sup>k</sup> | Х | | | At the disc | cretion of | the investig | ator, if clir | nically indic | cated, until | disease p | rogression | |
| Bone Scan/Imaging <sup>I</sup> | Х | | | | | ı | As clinical | ly indicate | d | | | |

#### Table 2Schedule of assessments for mGC patients (Phase I, Cohort 2) (cont.)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2- | -3 | Су | cle 4 onv | /ards | Safety<br>Follow-Up<br>Visit | Safety<br>Follow-Up <sup>3</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 6<br>months |
| Hematology <sup>m</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | Х | |
| Biochemistry <sup>o</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | Х | |
| Urinalysis <sup>p</sup> | Х | | As clinically indicated | | | | | Х | | | | |
| INR/aPTT | Х | P | As clinicall | y indicate | d, e.g. for | patients r | eceiving ar | nticoagulat | ion therap | ру | Х | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Xq | | | X <sup>q</sup> | Х | Х |
| PK/PD Samples (see Appendix 2) | | Х | | | Х | | | | | | | |
| Assessment of Patient<br>Hospitalizations and/or Hospital<br>Visits | | х | | | Х | | | Х | | | Х | |
| Administration of trastuzumab emtansine | | D 2 <sup>r</sup> | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Administration of capecitabine | | D 1–14 D 1–14 D 1–14 | | | | | | | | | | |
| Overall survival | Х | | X | | | | | Х | Х | | | |

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

- 1.NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within **14 days** prior to first study treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1) visit.
- 2.All patients will be followed up every 6 months (except for pregnancy which is every 3 months) until disease progression or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than disease progression will continue to undergo tumor assessments every 3-6 months.
- a)Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests.
- b)HER2-positivity is defined as IHC 3+ alone or IHC 2+ in combination with gene amplification by ISH. For mGC patients enrolled into Cohort 2, central confirmation of HER2 status is required.
- c)Limited symptom-directed physical examination.
- d)Height to be obtained at screening or at Cycle 1 Day 1 only.
- e)Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f)Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to fist study treatment.
- g)During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h)Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatment-related AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i)Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, and on Days 15–21, 30–42 and 9 weeks thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

- j)Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than disease progression, continued tumor assessments according to the protocol schedule of assessments is required.
- k)Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 4 months) as detailed in Section 4.4.1.4 of the protocol and in Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- I)An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed >28 days but ≤ 60 days prior to first study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- m)Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and WBC with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils).
- n)Assessments should be performed at screening, on Day 1, 8 and 15 of all cycles. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- o)Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, BUN/urea, creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN).
- p)Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.
- q)Serum β-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.
- r)Trastuzumab emtansine will be administered on Day 1 of each weekly cycle for all patients enrolled in Cohort 2 (A&B) except in the first cycle where trastzumab emtansine will be given on DAY 2 (to allow drug interaction assessment).

# Appendix 2 Pharmacokinetic Sampling for Phase I, Metastatic Breast and Gastric Cancer Patients

| | Trastuzumab<br>emtansine, total<br>trastuzumab and DM1<br>PK samples | Capecitabine and 5-FU<br>PK samples |
|---|---|---|
| Cycle 1 Day 1 | | |
| Pre capecitabine dose | | X |
| 30 min post capecitabine dosing | | X |
| 60 min post capecitabine dosing | | X |
| 1.5 hours post capecitabine dosing | | x |
| 2 hours post capecitabine dosing | | x |
| 2.5 hours post capecitabine dosing | | x |
| 4 hours post capecitabine dosing | | х |
| 6 hours post capecitabine dosing | | х |
| Cycle 1 Day 2 | | |
| Pre trastzumab emtansine dose | Х | |
| 15-30 minutes after end of trastuzumab emtansine infusion | х | |
| Cycle 2 Day 1 | | |
| Pre trastuzumab emtansine or capecitabine dose | X | x |
| 30 min post capecitabine dosing | | Х |
| 60 min post capecitabine dosing | | X |
| 1.5 hours post capecitabine dosing | | X |
| 15-30 min after end of trastuzumab emtansine infusion | х | |
| 2 hours post capecitabine dosing | | x |
| 2.5 hours post capecitabine dosing | | x |
| 4 hours post capecitabine dosing | | x |

# Appendix 2 Pharmacokinetic Sampling for Phase I, Metastatic Breast and Gastric Cancer Patients (cont.)

| | Trastuzumab<br>emtansine, total<br>trastuzumab and DM1<br>PK samples | Capecitabine and 5-FU<br>PK samples |
|---|---|---|
| 6 hours post capecitabine dosing | | х |
| Cycle 3 | | |
| Pre trastuzumab emtansine dose | x | |

PK = pharmacokinetic; 5-FU = 5-fluoruracil

Selected sections from the Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1,<sup>1</sup> are presented below, with slight modifications and the addition of explanatory text as needed for clarity.<sup>2</sup>

#### **Measurability of Tumor at Baseline**

#### **Definitions**

At baseline, tumor lesions/lymph nodes will be categorized as measurable or non-measurable as described below.

#### a. Measurable Tumor Lesions

**Tumor Lesions.** Tumor lesions must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size as follows:

- 10 mm by CT or magnetic resonance imaging (MRI) scan (CT/MRI scan slice thickness/interval no greater than 5 mm)
- 10-mm caliper measurement by clinical examination (lesions that cannot be accurately measured with calipers should be recorded as nonmeasurable)
- 20 mm by chest X-ray

**Malignant Lymph Nodes.** To be considered pathologically enlarged and measurable, a lymph node must be  $\geq 15$  mm in the short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and follow-up, only the short axis will be measured and followed. See also notes below on "Baseline Documentation of Target and Non-Target Lesions" for information on lymph node measurement.

<sup>&</sup>lt;sup>1</sup> Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (Version 1.1). Eur J Cancer 2009;45:228–47.

<sup>&</sup>lt;sup>2</sup> For consistency within this document, the section numbers and cross-references to other sections within the article have been deleted and minor formatting changes have been made.

#### b. Non-Measurable Tumor Lesions

Non-measurable tumor lesions encompass small lesions (longest diameter > 10 mm or pathological lymph nodes with short axis ≥ 10 but < 15 mm) as well as truly non-measurable lesions. Lesions considered truly non-measurable include leptomeningeal disease, ascites, pleural or pericardial effusion, inflammatory breast disease, lymphangitic involvement of skin or lung, peritoneal spread, and abdominal mass/abdominal organomegaly identified by physical examination that is not measurable by reproducible imaging techniques.

#### c. Special Considerations Regarding Lesion Measurability

Bone lesions, cystic lesions, and lesions previously treated with local therapy require particular comment, as outlined below.

#### Bone Lesions:

- Bone scan, PET scan, or plain films are not considered adequate imaging techniques for measuring bone lesions. However, these techniques can be used to confirm the presence or disappearance of bone lesions.
- Lytic bone lesions or mixed lytic-blastic lesions, with identifiable soft tissue components, that can be evaluated by cross-sectional imaging techniques such as CT or MRI can be considered as measurable lesions if the soft tissue component meets the definition of measurability described above.
- Blastic bone lesions are non-measurable.

#### Cystic Lesions:

- Lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor non-measurable) since they are, by definition, simple cysts.
- Cystic lesions thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of measurability described above. However, if non-cystic lesions are present in the same patient, these are preferred for selection as target lesions.

#### Lesions with Prior Local Treatment:

 Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion. Study protocols should detail the conditions under which such lesions would be considered measurable.

#### **Target Lesions: Specifications by Methods of Measurements**

#### a. Measurement of Lesions

All measurements should be recorded in metric notation, using calipers if clinically assessed. All baseline evaluations should be performed as close as possible to the treatment start and never more than 28 days before the beginning of the treatment.

#### b. Method of Assessment

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during the study. Imaging-based evaluation should always be the preferred option.

**Clinical Lesions.** Clinical lesions will only be considered measurable when they are superficial and ≥ 10 mm in diameter as assessed using calipers (e.g., skin nodules). For the case of skin lesions, documentation by color photography including a ruler to estimate the size of the lesion is suggested.

**Chest X-Ray.** Chest CT is preferred over chest X-ray, particularly when progression is an important endpoint, since CT is more sensitive than X-ray, particularly in identifying new lesions. However, lesions on chest X-ray may be considered measurable if they are clearly defined and surrounded by aerated lung.

**CT, MRI.** CT is the best currently available and reproducible method to measure lesions selected for response assessment. This guideline has defined measurability of lesions on CT scan based on the assumption that CT slice thickness is 5 mm or less. When CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness. MRI is also acceptable.

If prior to enrollment it is known that a patient is unable to undergo CT scans with IV contrast because of allergy or renal insufficiency, the decision as to whether a non-contrast CT or MRI (without IV contrast) will be used to evaluate the patient at baseline and during the study should be guided by the tumor type under investigation and the anatomic location of the disease. For patients who develop contraindications to contrast after baseline contrast CT is done, the decision as to whether non-contrast CT or MRI (enhanced or non-enhanced) will be performed should also be based on the tumor type and the anatomic location of the disease, and should be optimized to allow for comparison with the prior studies if possible. Each case should be discussed with the radiologist to determine if substitution of these other approaches is possible and, if not, the patient should be considered not evaluable from that point forward. Care must

be taken in measurement of target lesions on a different modality and interpretation of non-target disease or new lesions, since the same lesion may appear to have a different size using a new modality.

**Ultrasound.** Ultrasound is not useful in assessment of lesion size and should not be used as a method of measurement.

Endoscopy, Laparoscopy, Tumor Markers, Cytology, Histology. The utilization of these techniques for objective tumor evaluation cannot generally be advised.

#### **Tumor Response Evaluation**

#### **Assessment of Overall Tumor Burden and Measurable Disease**

To assess objective response or future progression, it is necessary to estimate the overall tumor burden at baseline and use this as a comparator for subsequent measurements. Measurable disease is defined by the presence of at least one measurable lesion, as detailed above.

#### **Baseline Documentation of Target and Non-Target Lesions**

When more than one measurable lesion is present at baseline, all lesions up to a maximum of five lesions total (and a maximum of two lesions per organ) representative of all involved organs should be identified as target lesions and will be recorded and measured at baseline. This means that, for instances in which patients have only one or two organ sites involved, a maximum of two lesions (one site) and four lesions (two sites), respectively, will be recorded. Other lesions (albeit measurable) in those organs will be recorded as non-measurable lesions (even if the size is > 10 mm by CT scan).

Target lesions should be selected on the basis of their size (lesions with the longest diameter) and be representative of all involved organs, but in addition should lend themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion does not lend itself to reproducible measurement, in which circumstance the next largest lesion that can be measured reproducibly should be selected.

Lymph nodes merit special mention since they are normal anatomical structures that may be visible by imaging even if not involved by tumor. As noted above, pathological nodes that are defined as measurable and may be identified as target lesions must meet the criterion of a short axis of  $\geq 15$  mm by CT scan. Only the short axis of these nodes will contribute to the baseline sum. The short axis of the node is the diameter normally used by radiologists

to judge if a node is involved by solid tumor. Nodal size is normally reported as two dimensions in the plane in which the image is obtained (for CT this is almost always the axial plane; for MRI the plane of acquisition may be axial, sagittal, or coronal). The smaller of these measures is the short axis. For example, an abdominal node that is reported as being 20 mm × 30 mm has a short axis of 20 mm and qualifies as a malignant, measurable node. In this example, 20 mm should be recorded as the node measurement. All other pathological nodes (those with short axis ≥ 10 mm but < 15 mm) should be considered non-target lesions. Nodes that have a short axis of < 10 mm are considered non-pathological and should not be recorded or followed.

A sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the baseline sum of diameters. If lymph nodes are to be included in the sum, then, as noted above, only the short axis is added into the sum. The baseline sum of diameters will be used as a reference to further characterize any objective tumor regression in the measurable dimension of the disease.

All other lesions (or sites of disease), including pathological lymph nodes, should be identified as non-target lesions and should also be recorded at baseline. Measurements are not required and these lesions should be followed as "present," "absent," or in rare cases "unequivocal progression."

In addition, it is possible to record multiple non-target lesions involving the same organ as a single item on the Case Report Form (CRF) (e.g., "multiple enlarged pelvic lymph nodes" or "multiple liver metastases").

#### Response Criteria

#### a. Evaluation of Target Lesions

This section provides the definitions of the criteria used to determine objective tumor response for target lesions.

- Complete response (CR): Disappearance of all target lesions
   Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.</li>
- Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters
- Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline

In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.

The appearance of one or more new lesions is also considered progression.

 Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study

#### b. Special Notes on the Assessment of Target Lesions

**Lymph Nodes.** Lymph nodes identified as target lesions should always have the actual short axis measurement recorded (measured in the same anatomical plane as the baseline examination), even if the nodes regress to < 10 mm on study. This means that when lymph nodes are included as target lesions, the sum of lesions may not be zero even if CR criteria are met, since a normal lymph node is defined as having a short axis of < 10 mm.

Target Lesions That Become too Small to Measure. During the study, all lesions (nodal and non-nodal) recorded at baseline should have their actual measurements recorded at each subsequent evaluation, even when very small (e.g., 2 mm). However, sometimes lesions or lymph nodes that are recorded as target lesions at baseline become so faint on CT scan that the radiologist may not feel comfortable assigning an exact measure and may report them as being too small to measure. When this occurs, it is important that a value be recorded on the CRF, as follows:

- If it is the opinion of the radiologist that the lesion has likely disappeared, the measurement should be recorded as 0 mm.
- If the lesion is believed to be present and is faintly seen but too small to measure, a default value of 5 mm should be assigned and below measuralble limit (BML) should be ticked. (Note: It is less likely that this rule will be used for lymph nodes since they usually have a definable size when normal and are frequently surrounded by fat such as in the retroperitoneum; however, if a lymph node is believed to be present and is faintly seen but too small to measure, a default value of 5 mm should be assigned in this circumstance as well and BML should also be ticked).

To reiterate, however, if the radiologist is able to provide an actual measure, that should be recorded, even if it is below 5 mm, and in that case BML should not be ticked.

**Lesions That Split or Coalesce on Treatment.** When non-nodal lesions fragment, the longest diameters of the fragmented portions should be added

together to calculate the target lesion sum. Similarly, as lesions coalesce, a plane between them may be maintained that would aid in obtaining maximal diameter measurements of each individual lesion. If the lesions have truly coalesced such that they are no longer separable, the vector of the longest diameter in this instance should be the maximum longest diameter for the coalesced lesion.

#### c. Evaluation of Non-Target Lesions

This section provides the definitions of the criteria used to determine the tumor response for the group of non-target lesions. While some non-target lesions may actually be measurable, they need not be measured and instead should be assessed only qualitatively at the time points specified in the protocol.

- Complete response (CR): Disappearance of all non-target lesions and (if applicable) normalization of tumor marker level
  - All lymph nodes must be non-pathological in size (< 10 mm short axis).
- Non-CR/Non-PD: Persistence of one or more non-target lesions and/or (if applicable) maintenance of tumor marker level above the normal limits
- Progressive disease (PD): Unequivocal progression of existing non-target lesions

The appearance of one or more new lesions is also considered progression.

#### d. Special Notes on Assessment of Progression of Non-Target Disease

When the Patient Also Has Measurable Disease. In this setting, to achieve unequivocal progression on the basis of the non-target disease, there must be an overall level of substantial worsening in non-target disease in a magnitude that, even in the presence of SD or PR in target disease, the overall tumor burden has increased sufficiently to merit discontinuation of therapy. A modest increase in the size of one or more non-target lesions is usually not sufficient to qualify for unequivocal progression status. The designation of overall progression solely on the basis of change in non-target disease in the face of SD or PR of target disease will therefore be extremely rare.

When the Patient Has Only Non-Measurable Disease. This circumstance arises in some Phase III trials when it is not a criterion of study entry to have measurable disease. The same general concepts apply here as noted above; however, in this instance there is no measurable disease assessment to factor into the interpretation of an increase in non-measurable disease burden. Because worsening in non-target disease cannot be easily quantified (by definition: if all lesions are truly non-measurable), a useful test that can be

applied when assessing patients for unequivocal progression is to consider if the increase in overall disease burden based on the change in non-measurable disease is comparable in magnitude to the increase that would be required to declare PD for measurable disease, that is, an increase in tumor burden representing an additional 73% increase in volume (which is equivalent to a 20% increase in diameter in a measurable lesion). Examples include an increase in a pleural effusion from "trace" to "large" or an increase in lymphangitic disease from localized to widespread, or may be described in protocols as "sufficient to require a change in therapy." If unequivocal progression is seen, the patient should be considered to have had overall PD at that point. While it would be ideal to have objective criteria to apply to non-measurable disease, the very nature of that disease makes it impossible to do so; therefore, the increase must be substantial.

#### e. New Lesions

The appearance of new malignant lesions denotes disease progression; therefore, some comments on detection of new lesions are important. There are no specific criteria for the identification of new radiographic lesions; however, the finding of a new lesion should be unequivocal, that is, not attributable to differences in scanning technique, change in imaging modality, or findings thought to represent something other than tumor (for example, some "new" bone lesions may be simply healing or flare of pre-existing lesions). This is particularly important when the patient's baseline lesions show partial or CR. For example, necrosis of a liver lesion may be reported on a CT scan report as a "new" cystic lesion, which it is not.

A lesion identified during the study in an anatomical location that was not scanned at baseline is considered a new lesion and will indicate disease progression.

If a new lesion is equivocal, for example because of its small size, continued therapy and follow-up evaluation will clarify if it represents truly new disease. If repeat scans confirm there is definitely a new lesion, then progression should be declared using the date of the initial scan.

#### **Evaluation of Response**

#### a. Time Point Response (Overall Response)

It is assumed that at each protocol-specified time point, a response assessment occurs. **Table 1** provides a summary of the overall response status calculation at each time point for patients who have measurable disease at baseline.

When patients have non-measurable (therefore non-target) disease only, **Table 2** is to be used.

Table 1 Time Point Response: Patients with Target Lesions (with or without Non-Target Lesions)

| Target Lesions | Non-Target Lesions | New Lesions | Overall Response |
|---|---|---|---|
| | CR | No | CR |
| CR | | | |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | NE |
| PD | Any | Yes or no | PD |
| Any | PD | Yes or no | PD |
| Any | Any | Yes | PD |

CR=complete response; NE=not evaluable; PD=progressive disease; PR=partial response; SD=stable disease.

Table 2 Time Point Response: Patients with Non-Target Lesions Only

| Non-Target Lesions | New Lesions | Overall Response |
|--------------------|-------------|------------------|
| | No | CR |
| CR | | |
| Non-CR/non-PD | No | Non-CR/non-PD a |
| Not all evaluated | No | NE |
| Unequivocal PD | Yes or no | PD |
| Any | Yes | PD |

CR = complete response; NE = not evaluable; PD = progressive disease.

<sup>&</sup>quot;Non-CR/non-PD" is preferred over "stable disease" for non-target disease since stable disease is increasingly used as an endpoint for assessment of efficacy in some trials; thus, assigning "stable disease" when no lesions can be measured is not advised.

#### b. Missing Assessments and Not Evaluable Designation

When no imaging/measurement is done at all at a particular time point, the patient is not evaluable at that time point. If only a subset of lesion measurements are made at an assessment, usually the case is also considered not evaluable at that time point, unless a convincing argument can be made that the contribution of the individual missing lesion(s) would not change the assigned time point response. This would be most likely to happen in the case of PD. For example, if a patient had a baseline sum of 50 mm with three measured lesions and during the study only two lesions were assessed, but those gave a sum of 80 mm, the patient will have achieved PD status, regardless of the contribution of the missing lesion.

If one or more target lesions were not assessed either because the scan was not done or the scan could not be assessed because of poor image quality or obstructed view, the response for target lesions should be "unable to assess" since the patient is not evaluable. Similarly, if one or more non-target lesions are not assessed, the response for non-target lesions should be "unable to assess" except where there is clear progression. Overall response would be "unable to assess" if either the target response or the non-target response is "unable to assess" except where this is clear evidence of progression, as this equates with the case being not evaluable at that time point.

#### c. Special Notes on Response Assessment

When nodal disease is included in the sum of target lesions and the nodes decrease to "normal" size (<10 mm), they may still have a measurement reported on scans. This measurement should be recorded even though the nodes are normal in order not to overstate progression should it be based on increase in size of the nodes. As noted earlier, this means that patients with CR may not have a total sum of "zero" on the CRF.

Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic deterioration." Every effort should be made to document objective progression even after discontinuation of treatment. Symptomatic deterioration is not a descriptor of an objective response; it is a reason for stopping study therapy. The objective response status of such patients is to be determined by evaluation of target and non-target disease as shown in **Table 1**, **Table 2**, **Table 3**.

Table 3 Best Overall Response When Confirmation Is Required

| Overall Response at First<br>Time Point | Overall Response at<br>Subsequent Time Point | Best Overall Response |
|---|---|---|
| | CR | CR |
| CR | | |
| CR | PR | SD, PD, or PR <sup>a</sup> |
| CR | SD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| CR | PD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| CR | NE | SD, provided minimum<br>duration for SD was met;<br>otherwise, NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| PR | NE | SD, provided minimum<br>duration for SD was met;<br>otherwise, NE |
| NE | NE | NE |

CR=complete response; NE=not evaluable; PD=progressive disease; PR=partial response; SD=stable disease.

<sup>&</sup>lt;sup>a</sup> If a CR is truly met at the first time point, any disease seen at a subsequent time point, even disease meeting PR criteria relative to baseline, qualifies as PD at that point (since disease must have reappeared after CR). Best response would depend on whether the minimum duration for SD was met. However, sometimes CR may be claimed when subsequent scans suggest small lesions were likely still present and in fact the patient had PR, not CR, at the first time point. Under these circumstances, the original CR should be changed to PR and the best response is PR.

For equivocal findings of progression (e.g., very small and uncertain new lesions; cystic changes or necrosis in existing lesions), treatment may continue until the next scheduled assessment. If at the next scheduled assessment, progression is confirmed, the date of progression should be the earlier date when progression was suspected.

In studies for which patients with advanced disease are eligible (i.e., primary disease still or partially present), the primary tumor should also be captured as a target or non-target lesion, as appropriate. This is to avoid an incorrect assessment of CR if the primary tumor is still present but not evaluated as a target or non-target lesion.

### Appendix 4 Instructions for Scans in the Event of Isotope Shortage

Two key suppliers of Tc-99m generators (Chalk River Reactor, Canada and High Flux Reactor, the Netherlands) are expected to close. eSupplies from other reactor sources will be unable to meet the expected world-wide patient-care needs. As a result, significant shortages of Tc-99m are expected, and the instructions listed below should be followed:

- ECHO will be the preferred imaging modality over MUGA scans to evaluate cardiac function.
- Tc-99m bone scans should be obtained as part of the baseline tumor assessment in all patients and should be repeated to confirm a CR or if progression of existing bone lesions and/or the development of new bone lesions is clinically suspected.
  - If a bone scan cannot be performed at baseline or if the investigator suspects that a bone scan may not be able to be repeated during the course of the study because of the Tc-99m shortage, the investigator may choose F-18 NaF or FDG-PET scan as an alternative.
- If bone lesions are selected as index non-target lesions, they must be apparent on baseline CT scans or other radiographic modalities (e.g., skeletal X-rays that can be repeated in subsequent tumor assessments).
   Additional scans may be obtained to follow clinically important bone lesions if not visualized on the chest, abdomen, or pelvic CT scan.

These measures are intended to ensure that the same method of assessment and the same imaging technique is used throughout the study for each patient. If there is a question regarding the choice of alternatives in the event that a standard bone scan cannot be obtained during screening and/or during the study, please contact the Medical Monitor.

# Appendix 5 New York Heart Association Classification of Functional Cardiac Capacity

| Class | |
|---|---|
| I | No limitation: Ordinary physical activity does not cause undue fatigue, dyspnea, or palpitation. |
| II | Slight limitation of physical activity: Such patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitations, dyspnea, or angina. |
| III | Marked limitation of physical activity: Although patients are comfortable at rest, less than ordinary physical activity will lead to symptoms. |
| IV | Inability to carry on physical activity without discomfort: Symptoms of congestive heart failure are present even at rest. With any physical activity, increased discomfort is experienced. |

From: Criteria Committee, New York Heart Association, Inc. Diseases of the heart and blood vessels. Nomenclature and criteria for diagnosis. 6th ed. Boston, Little, Brown and Co, 1964:114.

#### **PROTOCOL**

TITLE: PHASE I STUDY OF THE COMBINATION OF TRASTUZUMAB

EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED OR METASTATIC GASTRIC CANCER PATIENTS, FOLLOWED BY A RANDOMIZED, OPEN-LABEL PHASE II STUDY OF T-DM1 AND CAPECITABINE VERSUS T-DM1 ALONE IN HER2-

POSITIVE METASTATIC BREAST CANCER

PROTOCOL NUMBER: MO28230 VERSION NUMBER: 2

**EUDRACT NUMBER:** 2012-001547-46


MEDICAL MONITOR: MD

SPONSOR: F. Hoffmann-La Roche Ltd

DATE FINAL: Last date of signatures below

#### FINAL PROTOCOL APPROVAL




The information contained in this document, especially any unpublished data, is the property of F. Hoffmann-La Roche Ltd (or under its control) and therefore is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Ethics Committee or Institutional Review Board. It is understood that this information will not be disclosed to others without written authorization from Roche except to the extent necessary to obtain informed consent from persons to whom the drug may be administered.

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 2, 03 September 2013

#### **TABLE OF CONTENTS**

| PR | OTOCOL ACC | CEPTANCE FORM | 10 |
|---|---|---|---|
| PR | OTOCOL SYN | NOPSIS | 11 |
| 1. | BACKGROU | IND | 27 |
| | 1.1 | Background on Disease | 27 |
| | 1.1.1 | HER2-Positive Breast Cancer, Metastatic Breast Cancer | 27 |
| | 1.1.2 | HER2-Positive Locally Advanced or Metastatic Gastric Cancer | 28 |
| | 1.2 | Background on Study Drugs | 29 |
| | 1.2.1 | Trastuzumab Emtansine | 29 |
| | 1.2.1.1 | Study TDM3569g | 31 |
| | 1.2.1.2 | Study TDM4258g | 31 |
| | 1.2.1.3 | Study TDM4374g | 32 |
| | 1.2.1.4 | Study TDM4450g | 33 |
| | 1.2.1.5 | Study TDM4688g | 34 |
| | 1.2.1.6 | Phase III Study TDM4370g | 34 |
| | 1.2.1.7 | Pharmacokinetics | 35 |
| | 1.2.2 | Capecitabine | 37 |
| | 1.2.2.1 | Study BO18255: Capecitabine and Trastuzumab in mGC | 37 |
| | 1.2.3 | Preclinical Data of the Combination of Trastuzumab Emtansine and a Fluoropyrimidine | 38 |
| | 1.3 | Study Rationale and Risk-Benefit Assessment | 40 |
| | 1.3.1 | For mBC | 40 |
| | 1.3.2 | For mGC | 41 |
| 2. | OBJECTIVE | S | 41 |
| | 2.1 | Phase I: MTD Finding of Trastuzumab Emtansine and Capecitabine in mBC | 41 |
| | 2.1.1 | Primary Objective | 41 |
| | 2.1.2 | Secondary Objectives | 41 |
| | 2.2 | Randomized Phase II: Exploration of Efficacy and Safety in mBC | 42 |
| | 2.2.1 | Primary Objective | 42 |
| | 2.2.2 | Secondary Objectives | 42 |

| | 2.3 | Phase I: MTD Finding of Trastuzumab Emtansine and Capecitabine in MGC | 42 |
|---|---|---|---|
| | 2.3.1 | Primary Objective | 42 |
| | 2.3.2 | Secondary Objectives | 42 |
| 3. | STUDY DES | IGN | 42 |
| | 3.1 | Description of Study | 42 |
| | 3.1.1 | Overview of Study Design | 43 |
| | 3.1.1.1 | Overview of Phase I Design in Patients with mBC | 44 |
| | 3.1.1.2 | Overview of Phase II: Exploration of Efficacy and Safety in Patients with mBC | 47 |
| | 3.1.1.3 | Overview of Phase I Design in mGC Patients | 47 |
| | 3.1.1.4 | Number of Patients | 48 |
| | 3.1.1.5 | Number of Centers | 48 |
| | 3.1.2 | Steering Committee | 48 |
| | 3.1.3 | Independent Data Monitoring Committee | 49 |
| | 3.2 | End of Study | 49 |
| | 3.3 | Rationale for Study Design | 49 |
| | 3.3.1 | Rationale for Patient Group Selection | 49 |
| | 3.3.1.1 | Rationale for Phase I | 49 |
| | 3.3.1.2 | Rationale for Randomized Phase II | 50 |
| | 3.3.2 | Rationale for Investigational Medicinal Dose Selection | 51 |
| | 3.3.2.1 | In Patients with mBC | 51 |
| | 3.3.2.2 | In Patients with mGC | 51 |
| | 3.3.2.3 | Rationale for Duration of Treatment | 51 |
| | 3.3.3 | Pharmacokinetic Sampling Rationale | 52 |
| | 3.4 | Outcome Measures | 52 |
| | 3.4.1 | Phase I: mBC | 52 |
| | 3.4.1.1 | Primary Efficacy Outcome Measure | 52 |
| | 3.4.1.2 | Secondary Efficacy Outcome Measure | 52 |
| | 3.4.1.3 | Primary Safety Outcome Measure | 52 |
| | 3.4.1.4 | Secondary Safety Outcome Measures | 52 |
| | 3.4.1.5 | Pharmacokinetic Outcome Measures | 52 |
| | 3.4.2 | Randomized Phase II: Exploration of Efficacy and Safety in mBC | 53 |
| | 3.4.2.1 | Primary Efficacy Outcome Measure | 53 |

| | 3.4.2.2 | Secondary Efficacy Outcome Measures | <b>5</b> 3 |
|---|---|---|---|
| | 3.4.2.3 | Primary Safety Outcome Measure | <b>5</b> 3 |
| | 3.4.2.4 | Secondary Safety Outcome Measures | 53 |
| | 3.4.2.5 | Pharmacokinetic Outcome Measures | 54 |
| | 3.4.3 | Phase I: mGC | 54 |
| | 3.4.3.1 | Primary Efficacy Outcome Measure | 54 |
| | 3.4.3.2 | Secondary Efficacy Outcome Measure | 54 |
| | 3.4.3.3 | Primary Safety Outcome Measure | 54 |
| | 3.4.3.4 | Secondary Safety Outcome Measures | 54 |
| | 3.4.3.5 | Pharmacokinetic Outcome Measures | 54 |
| 4. | MATERIALS | AND METHODS | 55 |
| | 4.1 | Patients | 55 |
| | 4.1.1 | Patients with mBC | 55 |
| | 4.1.2 | mGC Patients | 55 |
| | 4.1.3 | Inclusion Criteria | 55 |
| | 4.1.3.1 | For Patients with mBC | 55 |
| | 4.1.3.2 | For Patients with mGC | <b>5</b> 6 |
| | 4.1.4 | Exclusion Criteria | 58 |
| | 4.1.4.1 | For Patients with mBC | 58 |
| | 4.1.4.2 | For Patients with mGC | 59 |
| | 4.1.5 | Patient Replacement Policy | 61 |
| | 4.2 | Method of Treatment Assignment | 61 |
| | 4.3 | Study Treatment | 61 |
| | 4.3.1 | Formulation, Packaging, and Handling | 61 |
| | 4.3.1.1 | Trastuzumab Emtansine | 61 |
| | 4.3.1.2 | Capecitabine | 62 |
| | 4.3.2 | Dosage and Administration | 63 |
| | 4.3.2.1 | For Patients with mBC | 63 |
| | 4.3.2.2 | For Patients with mGC | 64 |
| | 4.3.3 | Investigational Medicinal Product Accountability | 64 |
| | 4.3.4 | Post-trial Access to Extension Study | 64 |
| | 4.4 | Concomitant And Excluded Therapies | 65 |
| | 4.4.1 | Permitted Therapy | 65 |
| | 4.4.2 | Prohibited Therapy | 65 |

| | 4.5 | Study Assessments | 66 |
|---|---|---|---|
| | 4.5.1 | Description of Study Assessments | 66 |
| | 4.5.1.1 | Medical History and Demographic Data | 66 |
| | 4.5.1.2 | Vital Signs | 66 |
| | 4.5.1.3 | Physical Examinations | 67 |
| | 4.5.1.4 | Tumor and Response Evaluations | 67 |
| | 4.5.1.5 | Laboratory Assessments | 68 |
| | 4.5.1.6 | Electrocardiograms | 68 |
| | 4.5.1.7 | ECOG Performance Status | 68 |
| | 4.5.1.8 | ECHO/MUGA | 69 |
| | 4.5.2 | Timing of Study Assessments | 69 |
| | 4.5.2.1 | Screening and Pretreatment Assessments | 69 |
| | 4.5.2.2 | Assessments during Treatment | 70 |
| | 4.5.2.3 | Assessments at Study Completion/Early Termination Visit | 70 |
| | 4.5.2.4 | Follow-up Assessments | 71 |
| | 4.5.2.5 | Assessments at Unplanned Visits | 71 |
| | 4.6 | Patient, Study, and Site Discontinuation | 71 |
| | 4.6.1 | Patient Discontinuation | 71 |
| | 4.6.2 | Study Discontinuation | 72 |
| <b>5</b> . | ASSESSME | NT OF SAFETY | 72 |
| | 5.1 | Safety Plan | 72 |
| | 5.1.1 | Risks Associated with Trastuzumab Emtansine | 72 |
| | 5.1.1.1 | Cardiotoxicity | 72 |
| | 5.1.1.2 | Hematologic Toxicity (Thrombocytopenia) | 73 |
| | 5.1.1.3 | Hepatotoxicity | 73 |
| | 5.1.1.4 | Pulmonary Toxicity | 74 |
| | 5.1.1.5 | Infusion-related Reactions/Hypersensitivity | 75 |
| | 5.1.1.6 | Neurotoxicity | 75 |
| | 5.1.1.7 | Extravasation | 75 |
| | 5.1.1.8 | Trastuzumab Emtansine Dose Modification | 76 |
| | 5.1.2 | Risks Associated with Capecitabine | <b>7</b> 6 |
| | 5.1.3 | Risks Associated with Trastuzumab Emtansine and Capecitabine Combination | 76 |
| | 5.1.4 | Definition of Dose-limiting Toxicity | 77 |
| | 5.1.5 | Management of Specific Adverse Events | 78 |
| | | nsine—F. Hoffmann-La Roche Ltd<br>/ersion 2, 03 September 2013 | 5 |

| 5.1.5.1 | Trastuzumab Emtansine Dose Modification | 78 |
|---|---|---|
| 5.1 | .5.1.1 Trastuzumab Emtansine Dose Modification for Thrombocytopenia | 79 |
| 5.1 | .5.1.2 Trastuzumab Emtansine Dose Modification for Hepatotoxicity | 80 |
| 5.1<br>5.1 | <ul> <li>.5.1.2.1 Concurrent elevations of ALT/AST and bilirubin meeting Hy's Law laboratory criteria</li> <li>.5.1.2.2 Nodular regenerative hyperplasia (NRH)</li> <li>.5.1.2.3 Transaminase elevations or bilirubin elevation requiring dose adjustment</li> <li>.5.1.3 Trastuzumab Emtansine Dose</li> </ul> | 80 |
| 5.1 | Modification for Neurotoxicity | |
| 5.1 | .5.1.5 Trastuzumab Emtansine Dose Modification/Management for Infusion-related Reactions, Hypersensitivity Reactions | |
| 5.1 | .5.1.6 Trastuzumab Emtansine Dose Modification for Pulmonary Toxicity | |
| 5.1 | .5.1.7 Trastuzumab Emtansine Dose Modification for Extravasation | 84 |
| 5.1.5.2 | 2 Capecitabine Dosage Modification | 84 |
| 5.2 | Safety Parameters and Definitions | 85 |
| 5.2.1 | Adverse Events | 85 |
| 5.2.2 | Serious Adverse Events (Immediately Reportable to the Sponsor) | 86 |
| 5.2.3 | Protocol-defined Events of Special Interest/Non-Serious Expedited Adverse Events | |
| 5.2.4 | Pregnancy and Contraception | 87 |
| 5.3 | Methods and Timing for Capturing and Assessing Safety Parameters | 89 |
| 5.3.1 | Adverse Event Reporting Period | 89 |
| 5.3.2 | Eliciting Adverse Event Information | 90 |
| 5.3.3 | Assessment of Severity of Adverse Events | 90 |
| 5.3.4 | Assessment of Causality of Adverse Events | 91 |
| 5.3.5 | Procedures for Recording Adverse Events | 92 |
| 5.3.5.1 | Diagnosis <i>versus</i> Signs and Symptoms | 93 |
| 5.3.5.2 | 2 Adverse Events Occurring Secondary to<br>Other Events | 93 |
| 5.3.5.3 | Persistent or Recurrent Adverse Events | 93 |

| | 5.3.5.4 | Abnormal Laboratory Values | 94 |
|---|---|---|---|
| | 5.3.5.5 | Deaths | 94 |
| | 5.3.5.6 | Pre-Existing Medical Conditions | 94 |
| | 5.3.5.7 | Lack of Efficacy or Clinical Worsening | 95 |
| | 5.3.5.8 | Hospitalization or Prolonged Hospitalization | 95 |
| | 5.4 | Immediate Reporting Requirements from Investigator to the Sponsor | 95 |
| | 5.4.1 | Emergency Medical Contacts | 96 |
| | 5.4.2 | Reporting Requirements for Serious Adverse Events and Non-serious Adverse Events of Special Interest | 96 |
| | 5.4.3 | Reporting Requirements for Pregnancies | |
| | 5.4.3.1 | | |
| | 5.4.3.2 | | |
| | 5.4.3.3 | Abortions | 97 |
| | 5.4.3.4 | Congenital Anomalies/Birth Defects | 97 |
| | 5.5 | Follow-up of Patients after Adverse Events | 98 |
| | 5.5.1 | Investigator Follow-up | 98 |
| | 5.5.2 | Sponsor Follow-up | 98 |
| | 5.6 | Post-study Adverse Events | 98 |
| | 5.7 | Expedited Reporting to Health Authorities,<br>Investigators, Institutional Review Boards, and<br>Ethics Committees | 98 |
| 6. | STATISTICA | AL CONSIDERATIONS AND ANALYSIS PLAN | 99 |
| | 6.1 | Determination of Sample Size | 99 |
| | 6.2 | Summaries of Conduct of Study | 101 |
| | 6.3 | Summaries of Treatment Group Comparability | 102 |
| | 6.4 | Efficacy Analyses | 103 |
| | 6.4.1 | Primary Efficacy Endpoint | 103 |
| | 6.4.2 | Secondary Efficacy Endpoints | 104 |
| | 6.5 | Safety Analyses | 105 |
| | 6.6 | Pharmacodynamic Analyses | 107 |
| | 6.7 | Pharmacokinetic Analyses | 107 |
| | 6.8 | Exploratory Analyses | 108 |
| | 6.9 | Interim Analyses | 108 |

| 7. | DATA CO | DLLECTION AND MANAGEMENT | 109 |
|---|---|---|---|
| | 7.1 | Data Quality Assurance | 109 |
| | 7.2 | Electronic Case Report Forms | 109 |
| | 7.3 | Source Data Documentation | 110 |
| | 7.4 | Use of Computerized Systems | 110 |
| | 7.5 | Retention of Records | 110 |
| 8. | ETHICAL | CONSIDERATIONS | 111 |
| | 8.1 | Compliance with Laws and Regulations | 111 |
| | 8.2 | Informed Consent | 111 |
| | 8.3 | Institutional Review Board or Ethics Committee | 112 |
| | 8.4 | Confidentiality | 112 |
| | 8.5 | Financial Disclosure | 113 |
| 9. | | OCUMENTATION, MONITORING, AND TRATION | 113 |
| | 9.1 | Study Documentation | 113 |
| | 9.2 | Site Inspections | 113 |
| | 9.3 | Administrative Structure | 113 |
| | 9.4 | Publication of Data and Protection of Trade Secrets | 113 |
| | 9.5 | Protocol Amendments | 114 |
| 10. | REFERE | NCES | 115 |
| | | LIST OF TABLES | |
| Tab | le 1 | Cycle 1 Mean (s.d.) Pharmacokinetic Parameters for Trastuzumab Emtansine Following Trastuzumab Emtansine Administration Every 3 Weeks and Weekly in Study TDM3569g | 36 |
| Tab | le 2 | Dose Reduction for Trastuzumab Emtansine (Patients with mBC) | 79 |
| Tab | le 3 | Dose Reductions for Trastuzumab Emtansine (Patients with mGC) | |
| Tab | le 4 | Trastuzumab Emtansine Dose Modification: Total Serum Bilirubin | 81 |
| Table 5 | | Trastuzumab Emtansine Dose Modification: Serum ALT or AST | |
| Tab | | Adverse Event Severity Grading Scale | 91 |
| ıab | le 7 | Guidance for Causal Attribution of Adverse Event/Serious Adverse Event | 92 |
| Tab | le 8 | Sample Size Based on BOR | 100 |

#### **LIST OF FIGURES**

| Figure 1 | Molecular Structure of Trastuzumab Emtansine | 30 |
|---|---|---|
| Figure 2 | MMTV HER2 Fo5 Mammary Tumor Transplants | 39 |
| Figure 3 | Anti-tumor Activity of Trastuzumab Emtansine in | |
| | Combination with Capecitabine in NCI-N87 | 39 |
| Figure 4 | Overview of Study Design | |
| Figure 5 | Overview of Phase I Dose Finding Study Design | 45 |
| Figure 6 | Algorithm for Continuation and Discontinuation of | |
| | Trastuzumab Emtansine Based on Left Ventricular | |
| | Ejection Fraction Assessments in Patients | 83 |
| | LIST OF APPENDICES | |
| Appendix 1 | Schedule of Assessments | 119 |
| Appendix 2 | Pharmacokinetic Sampling for Phase I, Metastatic | |
| , трропал = | Breast and Gastric Cancer Patients | 128 |
| Appendix 3 | Response Evaluation Criteria in Solid Tumors | |
| | (RECIST): Modified Excerpt from Original Publication | 130 |
| Appendix 4 | Instructions for Scans in the Event of Isotope Shortage | 142 |
| p p o como | | |
| Appendix 5 | New York Heart Association Classification of | |
| | Functional Cardiac Capacity | 143 |
| Appendix 6 | ECOG Performance Status | 144 |
| , woodiidin U | EUUU I UHUHHUU Ulaluu | |
# PROTOCOL ACCEPTANCE FORM

TITLE: PHASE I STUDY OF THE COMBINATION OF TRASTUZUMAB EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED OR METASTATIC GASTRIC CANCER PATIENTS, FOLLOWED BY A RANDOMIZED, OPEN-LABEL PHASE II STUDY OF T-DM1 AND CAPECITABINE VERSUS T-DM1 ALONE IN HER2-

| OF T-DM1 AND CAPECITABINE VERSUS T-DM1 ALONE IN HER2-<br>POSITIVE METASTATIC BREAST CANCER | | |
|---|---|---|
| PROTOCOL NUMBER: | MO28230 | <b>VERSION NUMBER:</b> 2 |
| EUDRACT NUMBER: | 2012-001547-46 | |
| IND NUMBER | To be determined | |
| MEDICAL MONITOR: | | |
| SPONSOR: | F. Hoffmann-La Roche Ltd | |
| I agree to conduct the study in accordance with the current protocol. | | |
| Principal Investigator's Name ( | | |
| Principal Investigator's Signatu | ıre | Date |

Please return the signed original of this form {as instructed by XX [e.g., your local study monitor, the CRO]} [or] {to the contact provided below}. Please retain a copy for your study files.

{Name} {Address}

#### **PROTOCOL SYNOPSIS**

TITLE: PHASE I STUDY OF THE COMBINATION OF TRASTUZUMAB EMTANSINE
(T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST
CANCER AND HER2-POSITIVE LOCALLY ADVANCED OR METASTATIC
GASTRIC CANCER PATIENTS, FOLLOWED BY A RANDOMIZED, OPEN-LABEL
PHASE II STUDY OF T-DM1 AND CAPECITABINE VERSUS T-DM1 ALONE IN
HER2-POSITIVE METASTATIC BREAST CANCER


**EUDRACT NUMBER:** 2012-001547-46


PHASE: I/II

**INDICATION:** HER2-positive metastatic breast and locally advanced or metastatic

gastric cancer

SPONSOR: F. Hoffmann-La Roche Ltd

#### **Objectives**

# Phase I: Maximum Tolerated Dose Finding of Trastuzumab Emtansine and Capecitabine in Metastatic Breast Cancer

#### **Primary Objective**

 To determine the maximum tolerated dose (MTD) of the combination of trastuzumab emtansine and capecitabine in metastatic breast cancer (mBC) patients

### Secondary Objectives

- Pharmacokinetics (PK) of trastuzumab emtansine and metabolites and capecitabine
- Safety of the combination of trastuzumab emtansine and capecitabine
- Overall response rate (ORR)

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

#### **Primary Objective**

 To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine in mBC patients, as measured by ORR by Response Evaluation Criteria for Solid Tumors (RECIST) v.1.1 per investigator local assessment

#### Secondary Objectives

- Safety profile of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine
- To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine in mBC patients, as measured by:
  - Time to response (TTR)
  - Duration of response (DoR)
  - Time to progression (TTP)
  - Time to treatment failure (TTF)
  - · Progression-free survival (PFS)
  - Clinical benefit rate (CBR)
  - Overall survival (OS)

## Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

# Phase I: MTD Finding of Trastuzumab Emtansine and Capecitabine in Metastatic Gastric Cancer

#### Primary Objective

• To determine the MTD of the combination of trastuzumab emtansine and capecitabine in metastatic gastric cancer (mGC) patients

#### Secondary Objectives

- PK of trastuzumab emtansine and metabolites and capecitabine
- Safety of the combination of trastuzumab emtansine and capecitabine
- ORR

## **Study Design**

## **Description of Study**

This is an international, multicenter study.

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in human epidermal growth factor receptor 2 (HER2)-positive mBC and locally advanced or mGC patients using a Phase I design, followed by a randomized, open-label Phase II study to explore the efficacy and safety of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine in mBC patients. Results from the Phase I in mGC will be used as supporting information for future studies in the indication (see Figure 4 in the protocol).

#### Phase I: MTD Finding, Cohort 1: mBC

Cohort 1 will open first with a 3 plus 3 classical design. Cohort 1 will enroll patients with HER2-positive mBC. The dose tested of trastuzumab emtansine remains fixed at 3.6 mg/kg every 3 weeks (q3w) and 3 dose levels of capecitabine administered twice daily (bid) on Days 1 to 14 in cycles of 3 weeks will be tested. All patients will be treated until disease progression, intolerable toxicity, withdrawn consent, or death. All patients will be followed-up until withdrawn consent, death, or up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first.

#### Dose Levels Explored in Phase I, Cohort 1

Dose Level 1:  $750 \text{ mg/m}^2$  capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine Dose Level -1:  $700 \text{ mg/m}^2$  capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine Dose Level -2:  $650 \text{ mg/m}^2$  capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine The rules for determining the MTD are presented below.

If Dose Level 1 is proved too toxic (dose-limiting toxicity [DLT] > 1/3 or > 1/6), the dose will be de-escalated to one dose level below (Dose Level -1)

If Dose Level -1 is well tolerated (DLT  $\leq$  1/6), this dose will be considered the MTD and, following the independent Data Monitoring Committee (IDMC) agreement, will be further explored in the Randomized Phase II part of the study. If Dose Level -1 is too toxic (DLT  $\geq$ 1/6), the dose will be de-escalated to Dose Level -2.

If Dose Level -2 is well tolerated (DLT  $\leq$  1/6), this dose will be considered the MTD and, following iDMC approval, will be further explored in the Randomized Phase II part of the study. However, if Dose Level -2 is too toxic (DLT > 1/6), the combination may be considered unfeasible, recruitment will be closed and neither the Randomized Phase II nor mGC cohort will be opened. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the Steering Committee (SC).

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

Phase II will be conducted in mBC patients only. This part of the study will explore the efficacy and safety of the combination treatment of T-DM1 and capecitabine, at the established MTD, compared with T-DM1 alone in mBC patients.

Once the MTD in Cohort 1 is established, additional 117 HER2-positive mBC patients will be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to the Phase II part of the study; however, they will be followed-up until end of study (EOS).

Patients will be treated until disease progression/recurrence, intolerable toxicity, withdrawn consent, or death. If capecitabine needs to be discontinued for any reason, trastuzumab

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

196 Study MO28230

emtansine may continue, and the patient will be followed-up until EOS. In case of discontinuation of trastuzumab emtansine, patients will be followed-up until EOS.

All patients will be followed-up until withdrawn consent, death, or up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first.

## Phase I: MTD Finding, Cohort 2: mGC

Once the capecitabine MTD dose is established in Cohort 1, Cohort 2 will open, with a 3 plus 3 classical design to enroll HER2-positive mGC patients. Trastuzumab emtansine will be administered weekly at the dose of 2.4 mg/kg and capecitabine will start at the MTD dose defined in Cohort 1; capecitabine dose level may be de-escalated.

All patients will be treated until disease progression, intolerable toxicity, withdrawn consent, or death. All patients will be followed-up until withdrawn consent, death, or up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first.

The dose levels for capecitabine will be the same as described in Cohort 1, except for Dose Level 1, which will not be explored in mGC patients. Guidelines for dose escalation and deescalation are as follows:

If the MTD established in Cohort 1 is defined at Dose Level -1:

- This will be the starting dose in Cohort 2. If Dose Level -1 is well tolerated (DLT ≤ 1/6), this dose will be established as the MTD for mGC
- De-escalation: if Dose Level -1 is not tolerated in Cohort 2 (> 1/6 DLT), de-escalation will be to Dose Level -2

If the MTD established in Cohort 1 is defined at Dose Level -2:

- This will be the starting dose in Cohort 2. If Dose Level -2 is well tolerated (DLT ≤ 1/6), this dose will be established as the MTD for mGC
- De-escalation: if Dose Level -2 is not tolerated in Cohort 2 (> 1/6 DLT), the combination will be considered not feasible for mGC and Cohort 2 will be terminated. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the SC

# **Number of Patients**

Phase I, Cohort 1: mBC

A minimum of 6 and up to 18 patients will be enrolled.

Randomized Phase II: Exploration of Efficacy and Safety in mBC

Exploration of efficacy and safety in mBC will be based on 117 randomized patients in total.

Phase I, Cohort 2: mGC

A total of 3 to 12 patients will be enrolled.

## **Target Population**

Phase I, Cohort 1: mBC

HER2-positive mBC patients will be enrolled.

The patient's HER2 status will be considered positive if the local institution or reference lab reported Grade 3+ staining intensity (on a scale of 0 to 3) by means of immunohistochemistry (IHC) or fluorescent in situ hybridization (FISH).

The HER2 status will be retrospectively confirmed by IHC and/or FISH in a central laboratory using archival paraffin-embedded tumor tissue. Patients must have metastatic disease and/or locally recurrent disease not amenable to resection. Retrospective central confirmation will not impact the treatment decisions or primary endpoint of Phase I and will be used to validate efficacy analyses in Phase I.

Patients must have received at least one treatment regimen, which includes a chemotherapy agent and trastuzumab.

Randomized Phase II: Exploration of Efficacy and Safety in mBC

HER2-positive mBC patients will be randomized to one of the treatment groups receiving either the combination of trastuzumab emtansine (T-DM1) with capecitabine or T-DM1 alone. Retrospective central confirmation will be used to censor the efficacy population for the Randomized Phase II part of the study.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Patients must have received at least one treatment regimen, which includes a chemotherapy agent and trastuzumab.

#### Phase I, Cohort 2: mGC

HER2-positive locally advanced or mGC patients will be enrolled.

Patients must not have received prior chemotherapy for advanced/metastatic disease.

#### Inclusion Criteria:

#### For mBC Patients:

- 1. Age ≥ 18 years old.
- 2. Signed informed consent prior to any study specific procedure.
- 3. Able and willing to comply with protocol.
- 4. Negative serum pregnancy test for women of childbearing potential (including premenopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential.
- 5. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 6 months after the last dose of study treatment (see Section 5.2.4 in the protocol).
- 6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
- 7. Blood:
  - a) Platelet count > 100,000 cells/mm<sup>3</sup>
  - b) International normalized ratio (INR) < 1.5
  - c) Absolute neutrophil count (ANC) > 1,500 cells/mm<sup>3</sup>
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 8. Liver function:
  - a) Total bilirubin  $\leq 1.5 \times$  the upper limit of normal (ULN).
  - b) Serum glutamic oxaloacetic transaminase (SGOT)/aspartate transaminase (AST) and serum glutamic pyruvic transaminase (SGPT)/alanine transaminase (ALT) ≤ 2.5 × the ULN.
  - c) Alkaline phosphatase  $\leq 2.5 \times$  the ULN. Patients with hepatic and/or bone metastases: alkaline phosphatase  $\leq 5 \times$  the ULN.
  - d) Evidence of stable liver function during the month prior to enrollment with liver function tests' (LFTs) fluctuations not exceeding  $2.5 \times ULN$  (for AST, ALT) and  $1.5 \times ULN$  (for total bilirubin). Patients with bone metastases: AST and ALT  $\leq 5.0 \times ULN$ .
- 9. Renal function:
  - a) Serum creatinine of < 177 μmol/L or calculated creatinine clearance (CL)</li>
     > 50 mL/min. If urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate ≤ 1 g of protein/24 hours.
- 10. Cardiac function:
  - a) Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (ECHO) or multiple-gated acquisition (scan) (MUGA).
- 11. Histologically or cytologically confirmed breast cancer.
- 12. HER2-positive disease IHC 3+ or in situ hybridization (ISH) positive.
- 13. Tumor block or 15 slides available for retrospective central confirmation of HER2-positivity (central confirmation not necessary for enrollment).
- 14. mBC with at least one measurable lesion according to RECIST v.1.1.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- 15. Disease progression on at least one regimen containing trastuzumab and chemotherapy.
- 16. Patients must have recovered from previous treatments

#### For mGC Patients:

- 1. Age ≥ 18 years old.
- 2. Signed informed consent prior to any study specific procedure.
- 3. Able and willing to comply with protocol.
- 4. Negative serum pregnancy test for women of childbearing potential (including premenopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential.
- 5. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 6 months after the last dose of study treatment (see Section 5.2.4 in the protocol).
- 6. ECOG performance status of 0, 1, or 2.
- 7. Blood:
  - a) Platelet count > 100,000 cells/mm<sup>3</sup>.
  - b) INR < 1.5.
  - c) ANC > 1,500 cells/mm<sup>3</sup>.
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 8. Liver function:
  - a) Total bilirubin ≤ 1.5 × ULN.
  - b) SGOT/AST and SGPT/ALT ≤ 2.5 × the ULN.
  - c) Alkaline phosphatase ≤ 2.5 × the ULN. Patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × the ULN.
  - d) Evidence of stable liver function during the month prior to enrollment with LFTs fluctuations not exceeding 2.5 × ULN (for AST, ALT) and 1.5 × ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN.
- 9. Renal function:
  - a) Serum creatinine of < 177  $\mu$ mol/L or calculated creatinine CL > 50 mL/min. If urine dipstick for proteinuria is  $\geq$  2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate  $\leq$  1 g of protein/24 hours.
- 10. Cardiac function:
  - a) LVEF  $\geq$  50% by ECHO or MUGA.
- 11. Histologically or cytologically confirmed mGC or locally advanced gastric cancer.
- 12. HER2-positive tumor (primary tumor or metastatic lesion), defined as either IHC 3+ alone or IHC 2+ in combination with ISH+, prospectively confirmed by a Sponsor-designated central laboratory prior to enrollment. ISH positivity is defined as a ratio of ≥ 2.0 for the number of HER2 gene copies to the number of signals for CEP17.
  - a) Archival tumor samples obtained from primary or metastatic sites are acceptable.
  - b) Invasive tumor for central confirmation of HER2 status is required.
  - c) A formalin-fixed paraffin-embedded (FFPE) tissue block with at least 5 mm of invasive tumor for central confirmation is preferred. If FFPE tissue blocks (or partial block) are unavailable due to country or site regulations, a minimum of 8 freshly cut unstained slides MUST be available for central review of HER2 status.
- 13. Inoperable locally advanced or mGC.

#### **Exclusion Criteria:**

#### For mBC Patients:

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half-lives, whatever is longest.
  - b) Hormonal therapy within 14 days.
  - c) Trastuzumab within 21 days.
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received prior trastuzumab emtansine.
- 3. Prior treatment with capecitabine.
- 4. History of severe and unexpected reactions to fluoropyrimidine or with known hypersensitivity to fluorouracil.
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogues, such as brivudine.
  - b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product.
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>.
  - b) Epirubicin > 900 mg/m<sup>2</sup>.
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 28 days of first study drug administration.
- 9. Current peripheral neuropathy of Grade ≥ 3 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.4.0.
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above.
- 11. Current unstable ventricular arrhythmia requiring treatment.
- 12. History of symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] Classes II–IV).
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration.
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment.
- 15. Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy.
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease).
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment.
- Current pregnancy or lactation.
- 20. Current known active infection with human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C virus (HBV/HCV).
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV deoxyribonucleic acid (DNA) viral load per local guidelines.
- 21. Lapatinib ≤ 14 days before first study drug administration.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- 22. Previous radiotherapy for the treatment of unresectable, locally advanced/recurrent or mBC is not allowed if:
  - a) The last fraction of radiotherapy has been administered within 14 days prior to first study drug administration.
  - b) More than 25% of marrow-bearing bone has been irradiated.
  - c) The patient has not recovered from any resulting acute toxicity to Grade ≤ 1 prior to first study drug administration.
- 23. No signs and symptoms suggestive that the patient has dihydropyrimidine dehydrogenase (DPD) deficiency.

#### For mGC Patients:

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half-lives, whatever is longest.
  - b) Hormonal therapy within 14 days.
  - c) Trastuzumab within 21 days.
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received prior trastuzumab emtansine.
- 3. Prior treatment with capecitabine.
- 4. History of severe and unexpected reactions to fluoropyrimidine or with known hypersensitivity to fluorouracil.
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogues, such as brivudine.
  - b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product.
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>.
  - b) Epirubicin > 900 mg/m<sup>2</sup>.
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>.
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 28 days of first study drug administration.
- 9. Current peripheral neuropathy of Grade ≥ 3 per the NCI CTCAE, v4.0.
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above.
- 11. Current unstable ventricular arrhythmia requiring treatment.
- 12. History of symptomatic CHF (NYHA Classes II-IV).
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration.
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment.
- 15. Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy.
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- 20. Current known active infection with HIV, HBV, and/or HCV
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Previous chemotherapy for advanced/metastatic disease
  - a) Prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrollment into the study
- 22. No signs and symptoms suggestive that the patient has DPD deficiency
- 23. Lapatinib ≤ 14 days before first study drug administration

# Length of Study

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to be 2 years for Dose Finding and the Phase II/Exploration of Efficacy and Safety. All patients will be followed-up until withdrawn consent, death or up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first. In case Dose Level -2 is too toxic, the study may be terminated prematurely. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the SC.

#### **End of Study**

Last patient last visit (LPLV) as per definition is the last data collection point that can be either a clinic visit or a laboratory sample (see above length of study).

#### **Efficacy Outcome Measures**

Efficacy will be evaluated as per RECIST v.1.1.

- Best overall response (BOR) rate
- DoR
- TTR
- TTP
- TTF
- **PFS**
- CBR
- OS

### **Safety Outcome Measures**

- **DLT** assessment
- Incidence and severity by NCI CTCAE version 4.0 of adverse events (AEs), serious adverse events (SAEs), AEs that cause discontinuation from the study treatment, and AEs of special interest (AESIs)
- Fatal cases and causes of death
- Laboratory parameters
- LVEF
- Treatment exposure

# **Pharmacodynamic Outcome Measures**

Hospital visit parameters.

#### **Pharmacokinetic Outcome Measures**

PK will be evaluated during Phase I for both trastuzumab emtansine and capecitabine (see Appendix 1, Schedule of Assessment in the protocol). In addition, PK samples may be taken ad hoc, in case of SAE or unexpected toxicities, which may be suggestive of potential drug-drug interaction.

### **Investigational Medicinal Products**

#### For mBC Patients:

Trastuzumab emtansine will be administered q3w at a dose of 3.6 mg/kg intravenous (IV).

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 2, 03 September 2013

201

The total trastuzumab emtansine dose will be calculated based on the patient's weight on Day 1 of (or up to 3 days before) each cycle with no upper limit.

<u>Capecitabine</u> will be administered twice a day, orally for 14 days followed by a 7-day rest period at the Dose Levels 1 to -2 described in the 'Trial Design' section.

Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Rounding of capecitabine dose, based on 150 mg and 500 mg tablet strength will be allowed to the nearest target dose, based on patient body surface area (BSA).

#### For mGC Patients:

<u>Trastuzumab emtansine</u> will be administered on Day 1 of a weekly cycle at the dose of 2.4 mg/kg IV.

The total trastuzumab emtansine dose will be calculated based on the patient's weight on Day 1 of (or up to 3 days before) each cycle with no upper limit.

<u>Capecitabine</u> will be administered twice a day, orally for 14 days followed by a 7-day rest period at the Dose Levels -1 to -2 described in the 'Trial Design' section.

Capecitabine tablets should be swallowed with water within 30 minutes after a meal.

#### **Non-Investigational Medicinal Products**

Not applicable.

#### **Statistical Analysis**

The study will include 2 phases and 2 cohorts:

- Phase I, Cohort 1: mBC Dose Finding Cohort
- Randomized Phase II: Exploration of Efficacy and Safety in mBC
- Phase I, Cohort 2: mGC Dose Finding Cohort

There is no formal efficacy interim analysis. However, an independent data monitoring committee (IDMC) will advise whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 20 and 60 patients have received at least 3 cycles of treatment (Cycle 3 Day 1) in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II of the study or as requested.

Efficacy data will only be provided if required by the IDMC to estimate the risk-benefit balance for the patients. Further details on the function and logistics of the IDMC will be provided in the IDMC Charter.

Corresponding analyses as described in the protocol will be performed when all data for both study phases are collected and cleaned.

### Analysis of primary and secondary endpoints:

#### Analysis Populations:

### Phase I, Cohort 1: MTD Finding: mBC Patients

The main analysis population for DLT assessment is the DLT evaluable population, which is defined as all enrolled and treated patients who have not experienced any major protocol violations (including violations of the inclusion and exclusion criteria) and have completed Cycle 1.

The safety population (SP) will include all patients who received at least one dose of study medication during Phase I.

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

The main analysis population for the efficacy analysis will be the intent-to-treat (ITT) population, which will include all patients randomized in the Phase II part of the study. The per-protocol (PP) population will include all ITT patients who have at least one post-baseline tumor assessment during the Phase II part of the study and no major protocol violations, which will be defined in the statistical analysis plan (SAP).

The SP will include all patients who received at least one dose of study medication during the Randomized Phase II part of the study.

### Phase I, Cohort 2: MTD Finding, mGC Patients

The main analysis population for DLT assessment is the DLT evaluable population, which is defined as all enrolled and treated patients who have not experienced any major protocol

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Study MO28230

violation (including violation of the inclusion and exclusion criteria) and have completed Cycle 1.

The SP will include all patients who received at least one dose of study medication during Phase I.

### Efficacy Endpoints:

# Phase I, Cohort 1: MTD Finding, mBC

The primary objectives are reaching the MTD and establishing a safety profile.

ORR, as a main efficacy endpoint, will be assessed via BOR rate. The BOR is defined as the best response recorded from the date of enrollment until disease progression/recurrence, death, withdrawal of consent or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### Randomized Phase II: Exploration of Efficacy in mBC

The primary efficacy endpoint for the Phase II part of the study is the ORR, as assessed via BOR. The BOR is defined as the best response recorded from the start or randomization into the Phase II part of the study and until disease progression or recurrence, death, withdrawal of consent or EOS, whichever occurs first. To be assigned a status of partial response (PR) or complete response (CR), i.e., to be a responder, changes in tumor measurements must be confirmed by repeated assessments performed no less than 28 days after the response criteria are first met, i.e., patients need to have two consecutive assessments of PR or CR.

The emphasis of the exploratory Randomized Phase II part of the study will not be formal statistical hypothesis testing but the estimation of:

- The BOR rate with corresponding 95% confidence intervals (CIs) for each treatment group. The justification of the sample size is based on considerations regarding the width of 95% CIs for each treatment group estimate (precision of the corresponding estimate).
- The treatment effect (between treatment groups comparison) with corresponding 95% Cls

The number and proportions of responders and non-responders (based on BOR) together with the two-sided 95% Clopper-Pearson CIs will be presented for each treatment group. The difference in BOR between treatment groups will be displayed with associated 95% CIs using the Hauck-Anderson approach.

The secondary endpoints for the Phase II part of the study will be:

- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

Estimates for the survivor function of both treatment groups for TTR, DoR, TTP, TTF, PFS and OS will be obtained by using the Kaplan-Meier method. Hazard ratios and associated 95% CIs will be estimated from non-stratified and stratified (based on the stratification factor) Cox regression models.

Clinical benefit response will include patients whose best (confirmed) response was PR or CR, or stable disease (SD) that lasted at least 6 months. CBR will be summarized in a similar way to the primary efficacy endpoint, ORR, as assessed by BOR.

# Phase I, Cohort 2: MTD Finding: mGC

The primary objectives are reaching the MTD and establishing a safety profile. Efficacy endpoints will be analyzed in a similar way to Phase I, Cohort 1: mBC.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

#### Safety Endpoints:

#### Phase I, Cohort 1: MTD Finding: mBC

The number and proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

Safety parameters for this study part will be summarized by treatment dose. The summaries of AEs, SAEs, AEs that cause discontinuation from the study treatment, and AESIs (as described in Section 5) will be analyzed in a similar way to AEs in Phase II. The summaries will include all patients who received at least one dose of study medication.

The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry will be presented in shift tables of NCI-CTC grade at baseline *versus* worst grade during treatment for Phase I, Cohort 1, and overall.

LVEF will be summarized over time by means of mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications, and physical examinations will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### Randomized Phase II: Exploration of Safety in mBC

Safety endpoints will be summarized by treatment group.

Safety endpoints during the Randomized Phase II part of the study will be assessed via: total AEs, AEs Grade ≥ 3, SAEs, premature withdrawal from study medication, AESIs, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

The incidence of AEs and SAEs will be summarized according to the primary SOC and within each SOC, by MedDRA preferred term. Time to onset of the first episode of AESI will also be summarized via Kaplan-Meier method. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry will be presented in shift tables of NCI-CTC grade at baseline *versus* worst grade during treatment for the Randomized Phase II part of the study.

LVEF will be summarized over time by means of mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications, and physical examinations will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### Phase I, Cohort 2: MTD Finding: mGC

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

Safety parameters will be summarized in a similar way to Phase I, Cohort 1: mBC.

# Pharmacokinetic Analysis

The following PK parameters of trastuzumab emtansine and capecitabine (not limited to these listed) will be determined only in the Phase I part of the study in all patients who receive study treatment using either non-compartmental and/or population methods, if data allow:

• Serum concentrations of trastuzumab emtansine (conjugate) and total trastuzumab

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- Plasma concentrations of DM1, capecitabine and its active metabolite 5-fluorouracil (5-FU)
- Total exposure (area under the serum concentration-time curve [AUC])
- Maximum concentration (C<sub>max</sub>)
- CL
- Volume of distribution (V<sub>d</sub>)
- Terminal half-life (T<sub>1/2</sub>)

All PK parameters will be listed and tabulated by treatment dose and by Cohort. Descriptive summary statistics including arithmetic mean, geometric mean (e.g., AUC and  $C_{max}$ ), median, range, standard deviation (s.d.), and coefficient of variation will be presented for each Cohort. Nonlinear mixed effects modeling will be also used but details will be presented in the SAP.

#### **Exploratory Analyses**

For all patients a retrospective central confirmation of the HER2 status will be done. Further exploratory analysis for HER2-positive patients (based on central confirmation) will be done for selected endpoints, e.g. BOR and safety (AEs, SAEs, AEs with Grade ≥ 3, and AESIs).

Subgroup analysis for BOR, safety (AEs, SAEs, AEs with Grade  $\geq$  3, and AESIs) in the Randomized Phase II part of the study will be presented for both treatment groups: elderly *versus* younger patients, patients with ECOG 0–1 *versus* ECOG 2. More details will be presented in the SAP.

### Pharmacoeconomic Endpoint

The number of hospital visits, number of days admitted, and type of visits (emergency department *versus* inpatient care) will be collected and compared. The reason for admission (disease progression *versus* AE) will also be assessed.

#### **Determination of Sample Size**

#### Sample Size for Phase I: MTD Finding: mBC

This part will be based on a classical 3 plus 3 Phase I design. A minimum of 6 and up to 18 patients will be enrolled in Cohort 1. There is no formal sample size estimation for this part.

## Sample Size for Randomized Phase II: Exploration of Efficacy and Safety in mBC

Approximately 117 patients (78 patients in the combination of T-DM1 and capecitabine respective 39 patients in T-DM1 treatment group), including a 10% withdrawal rate, will be randomized with a 2:1 ratio to the combination of T-DM1 and capecitabine or T-DM1.

Point estimates and 95% Clopper-Pearson exact CIs are tabulated for a range of possible BOR outcomes for both treatment groups:

|--|

| Sample size based on BC | )R |
|---|---|
| N (T-DM1 and capecitabir | N (T-DM1 and capecitabine)* = 70 patients* |
| BOR rate [%] | 95% CI (within treatment group) [%] |
| 57.5 | (45.1–69.2) |
| 60.0 | (47.6–71.5) |
| 62.5 | (50.1–73.8) |
| 65.0 | (52.7–76.0) |
| 67.5 | (55.2–78.2) |
| N (T-DM1) = 35 patients* | |
| BOR rate [%] | 95% CI (within treatment group) [%] |
| 37.0 | (21.4–54.9) |
| 40.0 | (23.9–57.9) |
| 43.0 | (26.4–60.8) |
| 46.0 | (29.1–63.6) |
| 49.0 | (31.8–66.4) |
| * N = Number of patients w | ithout adjustment for withdrawal; CI = confidence interval |
| N (T-DM1 and capecitabine | e) / N (T-DM1) = 2 |

Expected BOR rate for patients who received trastuzumab emtansine of 43.6% (95% CI: 38.6% – 48.6%) was chosen based on previously published data for trastuzumab emtansine (see Section 6.1 of the main body of the protocol for reference).

The precision for the BOR estimate of the combination of T-DM1 and capecitabine is approximately 12%, e.g. BOR of 60%, 95% CI of (47.6%, 71.5%). Due to the lower sample size of the treatment group T-DM1, the corresponding precision for the BOR estimate is increased to 18%, e.g. BOR of 46%, 95% CI of (29.1%, 63.6%)

A 2:1 randomization will be applied to allow more patients being exposed to the combination of T-DM1 and capecitabine. This will enable a more thorough assessment of the corresponding safety profile.

# **Stratification Factors**

The following stratification factor will be implemented in the Randomized Phase II part of the study:

 Number of prior lines of treatment for metastatic disease (1 or >1; excluding singleagent hormones).

A treatment line is defined as any treatment regime given to patient from treatment initiation until confirmed disease progression.

## Sample Size for Phase I, Cohort 2: MTD Finding: mGC

This part will be based on a classical 3 plus 3 Phase I design. From 3 to 12 patients might be enrolled in Cohort 2. There is no formal sample size estimation for this part.

# **LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS**

| Abbreviation | Definition |
|------------------|------------------------------------------------|
| ADL | activities of daily living |
| AE | adverse event |
| AESI | adverse event of special interest |
| ADC | antibody-drug conjugate |
| ALT | alanine transaminase |
| ANC | absolute neutrophil count |
| aPTT | activated partial thromboplastin time |
| ARDS | acute respiratory distress syndrome |
| AST | aspartate transaminase |
| AUC | area under the serum concentration-time curve |
| BC | breast cancer |
| bid | twice daily |
| BML | below measurable limit |
| BOR | best overall response |
| BSA | body surface area |
| BUN | blood urea nitrogen |
| CBR | clinical benefit rate |
| CHF | congestive heart failure |
| CI | confidence interval |
| CL | clearance |
| C <sub>max</sub> | maximum concentration |
| CR | complete response |
| CRO | contract research organization |
| CSR | clinical study report |
| СТ | computed tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DLT | dose-limiting toxicity |
| DNA | deoxyribonucleic acid |
| DoR | duration of response |
| DPD | dihydropyrimidine dehydrogenase |
| 5-DFUR | 5'-deoxy-5-fluorouridine |
| 5-FU | 5-fluoruracil |
| EC | Ethics Committee |
| ECG | electrocardiogram |
| ECHO | echocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |

| EEA | European economic area |
|----------|-------------------------------------------------------------|
| EU | European Union |
| FDA | Food and Drug Administration |
| FFPE | formalin-fixed paraffin-embedded |
| FISH | fluorescence in situ hybridization |
| GC | gastric cancer |
| GCP | Good Clinical Practice |
| GEJ | gastroesophageal junction |
| HBV | hepatitis B virus |
| HCV | hepatitis C virus |
| HER2 | human epidermal growth factor receptor 2 |
| HIPAA | Health Insurance Portability and Accountability Act |
| HR | hazard ratio |
| HIV | human immunodeficiency virus |
| ICH | International Conference on Harmonisation |
| IDMC | independent data monitoring committee |
| IHC | immunohistochemistry |
| ILD | interstitial lung disease |
| IMP | investigational medicinal product |
| IND | Investigational New Drug (application) |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| ISH | in situ hybridization |
| ITT | intent-to-treat |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| IxRS | interactive voice/web recognition system |
| LC-MS/MS | liquid chromatography electrospray tandem mass spectrometry |
| LFT | liver function test |
| LPLV | last patient last visit |
| LVEF | left ventricular ejection fraction |
| mBC | metastatic breast cancer |
| mGC | metastatic gastric cancer |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | magnetic resonance imaging |
| MTD | maximum tolerated dose |
| MUGA | multiple-gated acquisition (scan) |
| N | number of patients |
| NCI | National Cancer Institute |
| NE | not evaluable |
| 1 | |

| NDU | nadular rapasarativa burarralasia |
|---|---|
| NRH<br>NYHA | nodular regenerative hyperplasia New York Heart Association |
| ORR | overall response rate |
| OS | overall survival |
| PD | pharmacodynamic/progressive disease |
| PET | positron emission tomography |
| PFS | progression-free survival |
| PK | pharmacokinetic |
| PP | per-protocol |
| PR | partial response |
| PVC | polyvinyl chloride |
| QTcF | heart rate-corrected QT interval using the Fridericia formula |
| q3w | every 3 weeks |
| qw | weekly |
| RECIST | Response Evaluation Criteria for Solid Tumors |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SGOT | serum glutamic oxaloacetic transaminase |
| SC | Steering Committee |
| s.d. | standard deviation |
| SD | stable disease |
| SDV | source data verification |
| SGPT | serum glutamic pyruvic transaminase |
| SOC | system-organ class |
| SP | safety population |
| SWFI | sterile water for injection |
| T <sub>1/2</sub> | terminal half-life |
| TTF | time to treatment failure |
| TTP | time to progression |
| TTR | time to response |
| ULN | upper limit of normal |
| $V_d$ | volume of distribution |
| WBC | white blood cells |
| WHO | World Health Organization |

# 1. BACKGROUND

# 1.1 BACKGROUND ON DISEASE

# 1.1.1 HER2-Positive Breast Cancer, Metastatic Breast Cancer

Breast cancer (BC) is the most common cancer in women worldwide, both in the developed and the developing world (WHO, World Health Statistics. 2011), with approximately 1.38 million new cases diagnosed in 2008. It is also the leading cause of cancer death in females, accounting for 458,400 deaths (14% of all cancer deaths) in 2008 (Jemal et al. 2011). Almost 100,000 of these BC-related deaths occurred in patients whose tumors overexpressed human epidermal growth factor receptor 2 (HER2) receptors. Metastatic breast cancer (mBC) is incurable, with the primary goal of treatment to extend life and palliate symptoms while preserving quality of life.

The HER tyrosine kinase receptor family is comprised of four receptors: HER1, HER2, HER3, and HER4. These receptors are important mediators of cell growth, survival, and differentiation (Sundaresan et al. 1999). Activation of HER receptors leads to receptor dimerization and cell signaling through the PI3-kinase/AKT pathway for promotion of tumor cell survival and through the mitogen-activated protein kinase pathway for cellular proliferation.

Overexpression of HER2 is observed in approximately 15–20% of human BCs. Several lines of scientific and clinical evidence support a direct role for HER2 overexpression in the aggressive growth and poor clinical outcomes associated with these tumors (Slamon et al. 1987). The development of trastuzumab in the 1990s provided women with HER2-overexpressing tumors with a markedly better outcome than was possible with chemotherapy alone. Increases in response rate, response duration, and progression-free survival (PFS) were associated with a 5-month survival advantage when trastuzumab was given in the first-line metastatic setting, as demonstrated in the initial Phase III trial (Slamon et al. 2001).

For patients with HER2-positive mBC, the combination of trastuzumab and a taxane is a globally accepted first-line treatment, based on the survival advantage demonstrated in two large pivotal trials (Slamon et al. 2001; Marty et al. 2005). However, virtually all patients with HER2-positive mBC develop progressive disease (PD) and require additional therapies. Importantly, such tumors continue to express high levels of HER2 (Spector et al. 2005), and neither the process of internalization nor the level of surface expression is altered when HER2 is bound by trastuzumab (Austin et al. 2004). HER2-directed combination therapy beyond progression for HER2-positive mBC is an accepted palliative treatment approach.

An accepted example of second-line therapy for HER2-positive mBC therapy is lapatinib in combination with capecitabine as a treatment for patients who have received trastuzumab and a taxane for advanced disease. In a Phase III trial involving patients with advanced HER2-positive BC previously treated

Study MO28230

with an anthracycline, a taxane, and trastuzumab, the addition of lapatinib to capecitabine resulted in an increased response rate (24% *versus* 14%) and time to disease progression (6.2 months *versus* 4.3 months) (Geyer et al. 2006).

Capecitabine (Xeloda®) in combination with docetaxel for treatment of patients with locally advanced or mBC after failure of cytotoxic chemotherapy. including an anthracycline was studied in a multicenter, randomized, controlled Phase III clinical trial (SO14999). In this trial, 255 patients were randomized to treatment with capecitabine (1,250 mg/m² twice daily [bid] for 2 weeks followed by a 1-week rest period) and docetaxel (75 mg/m<sup>2</sup> as a 1-hour intravenous [IV] infusion every 3 weeks [g3w]). A total of 256 patients were randomized to treatment with docetaxel alone (100 mg/m<sup>2</sup> as a 1-hour IV infusion q3w). Survival was superior in the capecitabine plus docetaxel combination arm (p = 0.0126). Median survival was 442 days (capecitabine plus docetaxel) versus 352 days (docetaxel alone). The overall objective response rates in the all-randomized population (investigator assessment) were 41.6% (capecitabine plus docetaxel) versus 29.7% (docetaxel alone); p = 0.0058. Time to progression (TTP) of disease or number of deaths was superior in the capecitabine plus docetaxel combination arm (p < 0.0001). The median TTP was 186 days (capecitabine plus docetaxel) versus 128 days (docetaxel alone).

Two multicenter Phase II clinical trials were conducted to determine the use of capecitabine monotherapy for treatment of patients with locally advanced or mBC after failure of a taxane and an anthracycline-containing chemotherapy regimen or for whom further anthracycline therapy is not indicated. In these trials, a total of 236 patients were treated with capecitabine (1,250 mg/m² bid for 2 weeks followed by 1-week rest period). The overall objective response rates (investigator assessment) were 20% (first trial) and 25% (second trial). The median TTP was 93 and 98 days. Median survival was 384 and 373 days (Blum et al. 1999; Blum et al. 2001).

# 1.1.2 HER2-Positive Locally Advanced or Metastatic Gastric Cancer

Gastric cancer (GC) remains one of the most common malignancies in the world with an estimated 989,600 new cases in 2008 (Jemal et al. 2011). GC also continues to be a deadly disease; it is the second leading cause of cancer-related death accounting for 738,000 deaths (9.7% of all cancer deaths) worldwide in 2008 (Ferlay et al. 2010). The only potentially curative treatment for GC is complete resection of localized disease. The overall 5-year survival for all cases, regardless of initial stage at diagnosis, is less than 25% (Catalano et al. 2005; Faivre et al. 1998; Parkin et al. 2005; Power et al. 2010). Among patients with localized disease who undergo curative surgery, approximately 40–60% will have disease recurrence. Patients with unresectable disease due to locally advanced growth or metastatic spread have the poorest prognosis, with an overall 5-year survival in the range of 3% to 15% (De Vivo et al. 2000; Ries et al. 2008; Power et al. 2010).

Whereas HER2 overexpression is associated with a poor prognosis in BC, the prognostic significance of HER2 overexpression in GC is not fully defined. Studies of HER2 positivity rates in GC have shown a broad variation of HER2 positivity ranging from 6.8% to 34.0% for immunohistochemistry (IHC) and 7.1% to 42.6% for fluorescence *in situ* hybridization (FISH) techniques (Hofmann et al. 2008; Tanner et al. 2005). In a recent study, HER2 positivity was shown in 17% of resected esophageal adenocarcinomas and was significantly associated with lower tumor grade, less invasiveness, fewer malignant nodes, and the presence of adjacent Barrett's esophagus (Yoon et al. 2012).

In the ToGA trial (study BO18255), a global, Phase III study of trastuzumab plus chemotherapy as first-line treatment for advanced HER2-positive GC, an overall HER2-positivity rate of 22.1% was observed (810/3667 evaluable samples), which is comparable to BC. A higher HER2-positivity rate was seen in adenocarcinoma of the gastroesophageal junction (GEJ) than in the stomach (33.2% *versus* 20.9%), and intestinal type GCs showed a significantly higher HER2-positivity rate than diffuse or mixed-type tumors (intestinal: 32.2%, diffuse: 6.1%, mixed: 20.4%; Albarello et al. 2011; Bang et al. 2010).

In the ToGA trial, the addition of trastuzumab to chemotherapy (capecitabine or fluorouracil combined with cisplatin) for the treatment of patients with HER2-positive (defined as IHC 3+ or FISH positive), inoperable, locally advanced or recurrent and/or metastatic adenocarcinoma of the stomach or GEJ resulted in an increase in the median overall survival (OS; 13.8 months *versus* 11.1 months, hazard ratio [HR] 0.74, p = 0.0046), objective response rate (47% *versus* 35%), PFS (6.7 *versus* 5.5 months), and TTP (7.1 *versus* 5.6 months) compared with chemotherapy alone (Bang et al. 2010).

# 1.2 BACKGROUND ON STUDY DRUGS

## 1.2.1 TRASTUZUMAB EMTANSINE

Trastuzumab emtansine (also known as T-DM1, see Figure 1) is a novel antibody-drug conjugate (ADC) that is specifically designed for the treatment of HER2-positive malignancies. Trastuzumab emtansine is composed of trastuzumab, a humanized monoclonal antibody directed against the extracellular region of HER2; an average of 3.5 molecules of DM1 (maytansinoid), an anti-microtubule agent derived from maytansine; and the thioether linker maleimidylmethyl cylcohexane-1-carboxylate, which is used to conjugate each molecule of DM1 to trastuzumab. DM1 is a highly potent drug synthesized from maytansinol that binds  $\beta$  tubulin to inhibit tubulin polymerization. It binds to tubulin competitively with vinca alkaloids, but is 20–100 times more potent than vincristine in its cytotoxic effect against tumor cell lines. Its parent molecule, maytansine, has been studied in approximately 800 cancer patients in the 1970s and 1980s, with responses seen in patients with breast and lung cancer (Junttila et al. 2011; Issell, Crooke 1978). However, because of its narrow therapeutic index and the observed

gastrointestinal toxicity of the free drug, it was not developed further as a therapeutic option (Cassady et al. 2004; Cabanillas et al. 1979).

Figure 1 Molecular Structure of Trastuzumab Emtansine



| | DM1<br>(derivative of maytansine) | Linker | rrastuzumar |
|--------|-----------------------------------|--------|-------------|
| MW: | 738 | 238 | ~150,000 |
| Ratio: | 3.5 | 3.5 | 1 |

DM1 = Derivative of Maytansine, a microtubule destabilizing agent MW = Molecular weight

Similar to trastuzumab, trastuzumab emtansine recognizes an epitope in the extracellular domain of HER2 and binds to HER2 with a similar affinity. Following antigen-specific binding of trastuzumab emtansine to HER2, the complex of receptor and ADC is internalized, whereupon DM1-containing catabolites are released into the cytosol following proteolytic cleavage of the antibody in lysosomes (Erickson et al. 2006). Binding of these DM1-containing species to  $\beta$ -tubulin inhibits tubulin polymerization resulting in cell death (Cassady et al. 2004).

In addition to targeting delivery of DM1 to HER2-overexpressing tumor cells, trastuzumab emtansine retains the anti-tumor activities of trastuzumab, including suppression of HER2 signaling pathways that confer a proliferative and survival advantage to cells, and the flagging of cells for destruction through antibody-dependent cell cytotoxicity (Junttila et al. 2011).

Completed and ongoing Phase I and II single-arm studies of trastuzumab emtansine have shown clinical activity. Furthermore, low levels of DM1 in systemic circulation supported the stability of the linker (Shen et al. ASCPT 2011). The randomized Phase II study TDM4450g described in Section 1.2.1.4 showed a significant improvement in PFS with a HR 0.59 (p = 0.0353) and a favorable safety profile. A Phase III study (TDM4370g) is underway comparing trastuzumab emtansine with HER2-targeted combination therapy (capecitabine and lapatinib) for patients with mBC who had received prior trastuzumab and taxane therapies.

Data from clinical trials of trastuzumab emtansine that are relevant to the design of the current trial are summarized below. Please refer to the trastuzumab emtansine Investigator's Brochure for further information on all of the completed and ongoing trastuzumab emtansine studies.

# 1.2.1.1 Study TDM3569g

Study TDM3569g was a Phase I, dose-escalation study that evaluated the safety and efficacy of trastuzumab emtansine as a single agent in 52 patients with HER2-positive mBC, whose disease progressed on a trastuzumab-containing chemotherapy regimen. The study was completed on 11 June 2009, with a total of 52 patients treated; 24 patients received trastuzumab emtansine q3w; 28 patients received trastuzumab emtansine on a weekly (qw) schedule.

On the q3w dosing schedule, dose-limiting toxicities of Grade 4 thrombocytopenia were seen in 2 of 3 patients treated at 4.8 mg/kg. Therefore, 3.6 mg/kg was determined to be the maximum tolerated dose (MTD) of trastuzumab emtansine given q3w, and the cohort was expanded to 15 patients. On the basis of these data, the recommended dose schedule for the Phase II studies was 3.6 mg/kg q3w. On the qw schedule, 2.4 mg/kg was identified as the MTD (Krop et al. 2008).

Treatment with trastuzumab emtansine was well tolerated, and toxicity was generally mild, reversible, and non-cumulative. No drug-related cardiac toxicity was noted.

Trastuzumab emtansine administration demonstrated considerable activity in this Phase I study. The confirmed overall response rate (ORR) in patients with measurable disease at the 3.6 mg/kg q3w schedule was 44% (4 of 9 patients), as assessed by investigators. The median PFS among the 15 patients receiving 3.6 mg/kg q3w was 10.4 months.

# 1.2.1.2 Study TDM4258g

Study TDM4258g was a Phase II study that evaluated the safety and efficacy of trastuzumab emtansine administered at a dose of 3.6 mg/kg (IV) q3w in patients with HER2-positive mBC who had progressed on previous HER2-directed therapy and conventional chemotherapy.

The primary objectives for this study were: 1) to assess the ORR (by independent radiologic review) associated with trastuzumab emtansine 3.6 mg/kg IV q3w, and 2) to characterize the safety and tolerability of trastuzumab emtansine at this dose.

The study was activated on 20 July 2007, and enrollment was completed (n = 112) on 31 July 2008. The final analysis of ORR was performed with a data cut-off date of 25 June 2009, 11 months after the last patient was enrolled. The reported ORR in all patients was 37.5% (95% confidence interval [CI]: 28.6%–46.6%) by investigator assessment and 25.9% (95% CI: 18.4%–34.4%) by Independent Review Board (IRB). The clinical benefit rate (CBR; defined as complete response [CR], partial response [PR], or stable

disease [SD] for >6 months) was 46.3% by investigator assessment and 39.3% by independent review. The median PFS was 4.6 months as assessed by both the investigators and the IRB. In the subset of patients whose archival primary tumors were retrospectively confirmed to be HER2-positive (74 of 95 patients with submitted tumor samples), the ORR was 33.8% by independent review and 47.3% based on investigator assessment.

The most common adverse events (AEs) (occurring in  $\geq$  20% of patients) were fatigue (65.2%), nausea (50.9%), headache (40.2%), epistaxis (35.7%), pyrexia (34.8%), constipation (30.4%), cough (27.7%), hypokalemia (26.8%), diarrhea (25.9%), vomiting (24.1%), arthralgia (22.3%), pain in extremity (22.3%), anemia (20.5%), and dyspnea (20.5%). Most of these AEs were Grade 1–2. The three most common Grade 3–4 AEs observed in this trial were hypokalemia (8.9%), thrombocytopenia (8.0%), and fatigue (4.5%). There was one reported Grade 5 event in a patient who died of respiratory failure attributed by the investigator to underlying disease. No Grade  $\geq$  3 left ventricular systolic dysfunction events (symptomatic congestive heart failure [CHF] and/or left ventricular ejection fraction [LVEF] of < 40%) were observed.

# 1.2.1.3 Study TDM4374g

Study TDM4374g was a Phase II, single-arm study of trastuzumab emtansine administered at 3.6 mg/kg by IV infusion q3w to patients with HER2-positive mBC. Patients must have received an anthracycline, trastuzumab, a taxane, lapatinib, and capecitabine given in the neoadjuvant, adjuvant, or metastatic setting or as treatment for locally advanced disease. Patients must have been treated with two HER2-directed therapies in the metastatic or locally advanced setting and have progressed on their most recent treatment.

The primary objectives of this study were: 1) to assess the ORR as assessed by an independent review using the modified Response Evaluation Criteria for Solid Tumors (RECIST) v. 1.0, and 2) to characterize the safety and tolerability of this trastuzumab emtansine regimen in the aforementioned patient population. The study was activated on 2 May 2008, and enrollment was complete on 2 April 2009. A total of 110 patients were enrolled and treated in the study.

An efficacy analysis (data cut-off date: 21 June 2010) with a median follow-up of 17.4 months demonstrated an ORR (complete and PR) of 34.5% (95% CI: 26.1%–43.9%; 38 of 110 patients) by independent review and 32.7% (95% CI: 24.1%–42.1%; 36 patients) by investigator assessment. The CBR was 48.2% by independent review and 46.4% by investigator assessment. The median duration of response (DoR) and PFS by independent review was 7.2 months and 6.9 months, respectively. In the subset of patients whose archival primary tumors were retrospectively confirmed to be HER2-positive (80 of 95 patients with submitted tumor samples), the ORR was 41.3% by independent review and 40.0% based on investigator assessment.

The most common AEs (occurring in  $\geq$  20% of patients) were fatigue (61.8%), thrombocytopenia (38.2%), nausea (37.3%), increased aspartate transaminase (AST, 26.4%), constipation (23.6%), pyrexia (22.7%), epistaxis

(22.7%), headache (21.8%), hypokalemia (20.9%), decreased appetite (20.9%), dry mouth (20.0%), and anemia (20.0%). Most of these AEs were Grade 1–2. Fifty-two patients (47.3%) experienced at least one Grade ≥ 3 AE, the most common being thrombocytopenia (9.1%) and fatigue (4.5%). Serious AEs (SAEs) were recorded by 28 patients (25.5%), the most common being cellulitis (3.6%), pyrexia (2.7%), and pneumonia (2.7%). One patient recorded a Grade 5 AE of hepatic dysfunction, which was recorded as possibly related to trastuzumab emtansine. The patient had pre-existing non-alcoholic fatty liver disease as well as multiple other comorbidities, including renal insufficiency.

# 1.2.1.4 Study TDM4450g

This was a randomized, multicenter, Phase II study of the efficacy and safety of trastuzumab emtansine *versus* trastuzumab plus docetaxel in patients with metastatic HER2-positive BC who had not received prior chemotherapy for metastatic disease. This study completed enrollment in December 2009 (n = 137). The primary objectives were to assess the efficacy of trastuzumab emtansine compared with the combination of trastuzumab and docetaxel, as measured by PFS based on investigator tumor assessments, and to characterize the safety of trastuzumab emtansine compared with the combination of trastuzumab and docetaxel in this population. Secondary endpoints included ORR, survival, and DoR.

The data cut-off date was 15 November 2010. Seventy patients were randomized to the control arm and 67 patients to the trastuzumab emtansine arm. The median duration of follow-up was 13.5 months for the control arm and 13.8 months for the trastuzumab emtansine arm.

As of 15 November 2010, the PFS was 14.2 months in the trastuzumab emtansine arm versus 9.2 months in the trastuzumab plus docetaxel arm. The HR for PFS was 0.594 (95% CI: 0.364-0.968; p = 0.0353). The ORR in the trastuzumab emtansine arm was 64.2% (95% CI: 51.8%-74.8%) compared with 58.0% (95% CI: 45.5%-69.2%) in the control arm (based on 69 evaluable patients). The CBR was 74.6% (95% CI: 63.2%-84.2%) in the trastuzumab emtansine arm versus 81.2% (95% CI: 70.7%-89.1%) in the trastuzumab plus docetaxel arm (based on 69 evaluable patients). Based on safety data analyzed at the data cut-off date, single-agent trastuzumab emtansine appears to have a favorable overall safety profile compared with trastuzumab and docetaxel in first-line mBC. The incidence of Grade ≥ 3 AEs in the control arm (89.4%; n = 66) was nearly twice that of trastuzumab emtansine (46.4%; n = 69). The rates of SAEs for both arms were similar (control arm 25.8% versus trastuzumab emtansine 18.8%). One patient in the trastuzumab emtansine group died as a result of an AE (sudden death). This patient was randomized to receive trastuzumab plus docetaxel but mistakenly received a single dose of 6 mg/kg trastuzumab emtansine instead of 6 mg/kg trastuzumab. One patient in the trastuzumab plus docetaxel group died due to cardiopulmonary failure. With respect to cardiotoxicity, based on local assessments of LVEF, trastuzumab emtansine was not associated with an increase in cardiotoxicity compared with trastuzumab plus docetaxel.

# 1.2.1.5 Study TDM4688g

The effect of trastuzumab emtansine (3.6 mg/kg q3w) on the QT interval in patients with HER2-positive recurrent locally advanced BC or mBC was evaluated in study TDM4688g, and had no meaningful effect on the corrected QT interval in these patients. At Cycle 1 Day 1, 15 minutes post-infusion, the baseline-adjusted mean heart rate-corrected QT interval using the Fridericia formula (QTcF) increased by 1.2 ms. By 60 minutes post-infusion, the baseline-adjusted mean QTcF interval decreased by 1.0 ms, and by Day 8 of Cycle 1, the baseline-adjusted mean QTcF interval decreased by 4.0 ms. By Cycle 3 Day 1, prior to trastuzumab emtansine infusion, the mean QTcF interval had reverted back to baseline. Following the third infusion of trastuzumab emtansine, the baseline-adjusted mean QTcF interval at both the 15 minute and the 60 minute post-infusion time points was increased by 4.7 ms. No patient exhibited a mean change in QTcF interval from baseline exceeding 30 ms at any of the protocol-specified time points.

The relationship between trastuzumab emtansine pharmacokinetic (PK) and electrocardiogram (ECG) data was also assessed. While there appears to be a trend between trastuzumab emtansine drug concentration and its effect on QT interval, at the observed concentration ranges of trastuzumab emtansine, DM1, and total trastuzumab, there is reasonable assurance that the true increase in mean baseline-adjusted average QTcF does not exceed 5 ms. Moreover, because trastuzumab emtansine, total trastuzumab, and DM1 achieve steady state levels by Cycle 3, the likelihood of progressively longer QTcF with repeated trastuzumab emtansine dosing is low.

In this study, an ORR of 25.5% (95% CI: 15.2%–38.5%) was assessed by the investigator; no independent review was performed in this study. The CBR was 39.2% (95% CI: 25.8%–53.1%), and the median PFS was 4.3 months (95% CI: 4.0–6.7).

# 1.2.1.6 Phase III Study TDM4370g

Roche is conducting a randomized, open-label Phase III trial (TDM4370g) of single-agent trastuzumab emtansine *versus* lapatinib and capecitabine in patients with HER2-positive locally advanced unresectable BC or mBC who have received a prior taxane and trastuzumab therapy and have documented disease progression. The study is ongoing, enrollment is completed, and 991 patients have been enrolled.

Patients are randomized in a 1:1 ratio to trastuzumab emtansine or capecitabine plus lapatinib.

Trastuzumab emtansine is administered at 3.6 mg/kg IV q3w. The control arm treatment is capecitabine at 1,000 mg/m² as oral doses bid on Days 1–14 of a q3w cycle plus oral lapatinib 1,250 mg/day given as continuous dosing. Study treatment is discontinued based on disease progression (as assessed by the investigator), unmanageable toxicity, or study termination by Roche/Genentech.

Study MO28230

This study of trastuzumab emtansine, met both primary efficacy endpoints of PFS by independent review and OS in patients with mBC previously treated with a taxane and trastuzumab (HERCEPTIN).

PFS and OS are investigated as co-primary endpoints in this study with PFS based on modified RECIST (Therasse et al. 2000) and conducted by the IRB. An additional tumor assessment of PFS is performed after investigator-documented disease progression. Furthermore ORR, DoR, and CBR are included, on the basis of both investigator and independent review of tumor assessments, as key secondary endpoints.

Patients in the trastuzumab emtansine arm had a median PFS of 9.6 months *versus* 6.4 months for patients in the control arm of lapatinib + capecitabine (HR = 0.65; 95% CI: 0.55–0.77; p < 0.001, log-rank test). Patients in the trastuzumab emtansine arm had a median OS of 30.9 months *versus* 25.1 months for patients in the control arm of lapatinib + capecitabine (HR = 0.68; 95% CI: 0.55–0.85; p < 0.001, log-rank test). The ORR in the trastuzumab emtansine arm was 43.6% (95% CI: 38.6%–48.6%) compared with 30.8% (95% CI: 26.3%–35.7%) in the control arm (based on 786 evaluable patients). Based on safety data analyzed at the data cut-off date, single-agent trastuzumab emtansine appears to have a favorable overall safety profile compared with lapatinib and capecitabine in mBC. The incidence of Grade  $\geq$  3 AEs in the control arm (56.9%; n = 488) was 278; that of trastuzumab emtansine (40.8%; n = 490) was 200. The rates of SAEs for both arms were similar (control arm 18% *versus* trastuzumab emtansine 15.5%).

It was concluded that overall, there is no concern regarding the clinical safety of trastuzumab emtansine for the patient population that was studied, based on the currently available data (Verma et al. 2012).

#### 1.2.1.7 Pharmacokinetics

The PK of trastuzumab emtansine and its analytes (total trastuzumab and DM1) were characterized in one Phase I study (TDM3569g) and three Phase II studies (TDM4258g, TDM4374g, and TDM4688g).

For study TDM3569g, the final PK parameter estimates based on non-compartmental PK analysis for q3w and qw regimens of trastuzumab emtansine administration are presented in Table 1.

Table 1 Cycle 1 Mean (s.d.) Pharmacokinetic Parameters for Trastuzumab Emtansine Following Trastuzumab Emtansine Administration Every 3 Weeks and Weekly in Study TDM3569g

| Dose | No. of | C <sub>max</sub> | AUC <sub>inf</sub> | T <sub>1/2</sub> | V <sub>d</sub> | CL |
|---|---|---|---|---|---|---|
| (mg/kg) | Patients | (µg/mL) | (day μg/mL) | (day) | (mL/kg) | (mL/day/kg) |
| Every 3 Week | Dosing | | | | | |
| 0.3 | 3 | 9.6 (1.7) | 14.5 (3.4) | 1.3 (0.2) | 35.7 (7.5) | 21.1 (4.5) |
| 0.6 | 1 | 13.3 | 24.5 | 1.3 | 43.8 | 24.5 |
| 1.2 | 1 | 20.3 | 42.9 | 1.3 | 51.8 | 27.8 |
| 2.4 | 1 | 76.3 | 330.0 | 2.2 | 30.7 | 7.2 |
| 3.6 | 15 | 76.2 (19.1) | 300.3 (65.8) | 3.1 (0.7) | 58.4 (12.4) | 12.7 (3.6) |
| 4.8 | 3 | 130.3 (7.8) | 673.0 (12.2) | 4.1 (0.7) | 41.2 (6.2) | 7.1 (0.1) |
| Weekly Dosing | g | | | | | |
| 1.2 | 3 | 29.6 (5.7) | 76.2 (10.4) | 2.3 (0.6) | 47.5 (6.0) | 15.9 (2.4) |
| 1.6 | 3 | 34.3 (4.8) | 130.3 (39.7) | 3.4 (0.8) | 59.8 (16.6) | 13.0 (3.4) |
| 2.0 | 3 | 48.0 (9.6) | 175.0 (41.0) | 3.1 (0.3) | 51.0 (8.1) | 11.8 (2.4) |
| 2.4 | 16 | 54.8 (12.6) | 198.5 (54.5) | 3.3 (1.1) | 55.4 (13.0) | 13.1 (4.1) |
| 2.9 | 3 | 78.1 (33.9) | 212.0 (39.0) | 2.9 (0.5) | 57.7 (2.2) | 14.0 (2.6) |

AUC<sub>inf</sub> = area under the serum concentration-time curve from time 0 extrapolated to infinity;  $C_{max}$  = maximum serum concentration; CL = clearance; s.d. = standard deviation;  $T_{1/2}$  = terminal half-life;  $V_{d}$  = volume of distribution.

Dose intensity, defined as percentage of the planned trastuzumab emtansine dose that was actually received, was higher with the 3.6 mg/kg q3w regimen (median 99.7%, range 88%–106%) than with the 2.4 mg/kg qw schedule (median 82%, range 54%–101%). However, since the PK of trastuzumab emtansine is linear at doses ≥ 2.4 mg/kg, an almost 2-fold higher cumulative dose can be administered within a q3w cycle with a 2.4 mg/kg qw regimen compared with 3.6 mg/kg q3w (Krop et al. 2009, Krop et al. 2010).

Based on a population PK analysis, trastuzumab emtansine has a consistent PK profile with low inter-individual variability (21%–48%) in PK parameters among patients with mBC. Greater baseline tumor burden and lower serum albumin levels, potential indicators of disease severity, resulted in small increases (< 13%) in trastuzumab emtansine clearance (CL). However, trastuzumab emtansine PK was not affected by baseline residual trastuzumab (from prior treatment) or by differences in serum concentrations of HER2 extracellular domain (Gupta et al. 2011).

An aggregate PK assessment of trastuzumab emtansine was performed with samples from studies TDM3569g, TDM4258g, TDM4374g, and TDM4688g (Girish et al. 2012; Igawa et al. 2012). PK parameters for trastuzumab emtansine, total trastuzumab, and DM1 were consistent across the four studies at Cycle 1 and steady state. Trastuzumab emtansine PK was not affected by residual trastuzumab from prior therapy or circulating extracellular domain of HER2. No significant correlations were observed between trastuzumab emtansine exposure and efficacy, thrombocytopenia, or

increased concentrations of transaminases. Across the four studies, the incidence of anti-therapeutic antibodies to trastuzumab emtansine was low and detected in 4.5% (13/286) of evaluable patients receiving trastuzumab emtansine q3w.

The PK profile (i.e., maximum concentration  $[C_{max}]$ , area under the serum concentration-time curve [AUC], terminal half-life  $[T_{1/2}]$ , apparent volume of distribution at steady state  $[V_{ss}]$ , and CL) of single-agent trastuzumab emtansine (3.6 mg/kg q3w) is predictable, well characterized, and unaffected by circulating levels of HER2 extracellular domain or residual trastuzumab. Trastuzumab emtansine exposure does not correlate with clinical responses or key AEs. Weekly administration of trastuzumab emtansine in study TDM3568g at a dose of 2.4 mg/kg showed consistent PK data with the q3w dosing schedule (Krop et al. 2008).

# 1.2.2 CAPECITABINE

Capecitabine (Xeloda<sup>®</sup>) is a fluoropyrimidine carbamate with antineoplastic activity. It is an orally administered systemic prodrug of 5'-deoxy-5-fluorouridine (5'-DFUR), which is converted to 5-fluorouracil (5-FU) in the tumor, where it inhibits DNA synthesis and slows down tumor tissue growth. It has been evaluated in clinical trials in combination with docetaxel and as monotherapy in BC (Geyer et al. 2006; Wardley et al. 2006; von Minckwitz et al. 2011). Please see the national Xeloda<sup>®</sup> prescribing information or Investigator brochure for more information.

# 1.2.2.1 Study BO18255: Capecitabine and Trastuzumab in mGC

Recently, a global Phase III study (ToGA trial, BO18255) of trastuzumab plus chemotherapy as first-line treatment for advanced HER2-positive GC was conducted in 584 patients previously untreated for HER2-positive inoperable locally advanced or recurrent and/or metastatic adenocarcinoma of the stomach or GEJ. Patients received either capecitabine or fluorouracil combined with cisplatin or the same chemotherapy in combination with trastuzumab. The primary study endpoint was OS, defined as the time from the date of randomization to the date of death from any cause. At the time of the analysis a total of 349 randomized patients had died: 182/290 patients (62.8%) in the control arm and 167/294 patients (56.8%) in the treatment arm. The majority of the deaths were due to events related to the underlying cancer (Bang et al. 2010).

Most patients enrolled in the study were male (76%); 52.9% were Asian and 37.7% were white. The primary tumor site was the stomach for 81.8% of patients, with the others having GEJ tumors. The addition of trastuzumab to chemotherapy resulted in an increase in median OS from 11.1 months to 13.8 months (HR 0.74, p = 0.0046). Objective response rate (47% *versus* 35%), PFS (6.7 *versus* 5.5 months), and TTP (7.1 *versus* 5.6 months) were also significantly increased with the addition of trastuzumab to chemotherapy compared with chemotherapy alone.

With regard to OS, a treatment effect could not be excluded in any predefined subgroup, including primary tumor site, histologic subtype, method of determining HER2-positivity, performance status, chemotherapy regimen, age, gender, and region of enrollment. A multivariate analysis for OS showed a consistent result, with an adjusted HR of 0.72 (p = 0.0036); variables found to influence primary outcome included Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1 *versus* 2), prior gastrectomy, and Asian region of enrollment (data on file). A multivariate analysis of OS for patients enrolled in Japan, from which the bulk of Asian patients were enrolled, demonstrated a HR of 0.68. This was consistent with the overall study results (Sawaki et al. 2012).

A pre-planned subgroup analysis by IHC score indicated that positive treatment effects are greater in tumors with higher levels of HER2 expression. Among patients whose tumors had these higher levels of HER2 expression, the median OS was 11.8 months versus 16 months (HR = 0.65; 95% CI: 0.51–0.83) and median PFS was 5.5 months versus 7.6 months (HR = 0.64; 95 % CI: 0.51–0.79) for chemotherapy versus chemotherapy plus trastuzumab respectively. For OS, the HR was 0.75 (95% CI: 0.51–1.11) in the IHC 2 + /FISH + group and 0.58 (95% CI: 0.41–0.81) in the IHC 3+/FISH+ group (Bang et al. 2010).

The addition of trastuzumab to chemotherapy did not result in an increased incidence of severe (Grade 3–4) or fatal (Grade 5) AEs. There were no additional significant safety issues with trastuzumab used in the treatment of advanced GC over and above those observed when it was used to BC. Taken together, the results of the ToGA trial (BO18255) not only demonstrate the role of HER2 suppression in the treatment of HER2-positive GC but also show that HER2-directed therapies can be added to conventional chemotherapy regimens without substantial increases in toxic side effects.

# 1.2.3 PRECLINICAL DATA OF THE COMBINATION OF TRASTUZUMAB EMTANSINE AND A FLUOROPYRIMIDINE

In BC preclinical models an additive anti-tumor activity was observed with combinations of trastuzumab emtansine and 5-FU (see Figure 2, [Lewis Phillips et al. 2008]). In GC models a similar additive effect was observed with trastuzumab emtansine and capecitabine (see Figure 3, [data on file]).

Figure 2 MMTV HER2 Fo5 Mammary Tumor Transplants



T-DM1 = trastuzumab emtansine; 5-FU = 5-fluoruracil

Figure 3 Anti-tumor Activity of Trastuzumab Emtansine in Combination with Capecitabine in NCI-N87



T-DM1 = trastuzumab emtansine; 5-FU = 5-fluoruracil

# 1.3 STUDY RATIONALE AND RISK-BENEFIT ASSESSMENT

# 1.3.1 FOR MBC

At present, mBC remains an incurable disease. The primary goal of treatment is maximizing the patient's survival and quality of life.

HER2-positive breast tumors have shown to benefit from anti-HER2 therapy. Regimens using the combination of anti-HER2 agents and chemotherapy have demonstrated higher efficacy than single-agent therapy. As a consequence several different combination therapies have been approved for HER2-positive mBC treatment in most countries and are considered the current standard of care.

The combination of capecitabine with anti-HER2 therapies has demonstrated to be beneficial for patients with mBC. The combination of capecitabine and lapatinib is approved in the United States since March 2007 for the treatment of patients with HER2-positive mBC who have previously received an anthracycline, a taxane, and trastuzumab. In June 2008, the European Commission granted conditional marketing authorization for lapatinib in combination with capecitabine for the treatment of patients with HER2-positive advanced or mBC who have previously received and progressed on an anthracycline, a taxane, and trastuzumab in the metastatic setting. The combination of capecitabine and trastuzumab has demonstrated significant efficacy benefit when compared with capecitabine alone (von Minckwitz et al. 2011).

In study TDM4450g, trastuzumab emtansine as a single agent showed a significant increase in PFS compared with the current standard of care of trastuzumab and a taxane (see Section 1.2.1.4), together with a favorable safety profile.

The Phase III, TDM4370g trial met its co-primary endpoint of improving PFS (by IRB) and OS compared with those who received the combination of lapatinib and capecitabine (see Section 1.2.1.6).

Based on the mentioned studies, the combination of trastuzumab emtansine and capecitabine could provide the potential for enhanced anti-tumor efficacy in mBC, compared with single-agent trastuzumab emtansine or trastuzumab in combination with chemotherapy.

Furthermore, preclinical data suggest that the combination of trastuzumab emtansine and capecitabine has an additive effect (see Section 1.2.3).

Approximately 2,000 patients with BC have been treated in trastuzumab emtansine clinical trials with an acceptable safety profile and a positive risk-benefit ratio. A broad development program is in place to seek approval for indications for mBC. Capecitabine in combination with anti-HER2 agent is a proven efficacious regimen with a well-established safety profile in mBC. Trastuzumab emtansine and capecitabine have no known significant overlapping toxicities. As a part of the Phase I conduct, regular teleconference calls with the investigators will be held to discuss the study treatment risk-

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 2, 03 September 2013 benefit profile for each patient. An IDMC will be established with the main responsibility to assess the risk-benefit for the Phase II part of the study. Therefore, exploring the benefit of combination therapy of trastuzumab emtansine and capecitabine in patients with mBC seems justified.

## 1.3.2 FOR MGC

As for mBC, the primary goal of treatment for metastatic gastric cancer (mGC) is the maximizing of the patient's survival and quality of life.

HER2-positive gastric tumors have shown to benefit from anti-HER2 therapy. Regimens using the combination of anti-HER2 agents and chemotherapy have demonstrated higher efficacy than single-agent therapy. As a consequence several different combination therapies have been approved for HER2-positive mGC treatment in most countries and are considered the current standard of care.

In HER2-positive mGC, the ToGA study (BO18255) has proven that the combination of chemotherapy and trastuzumab significantly improves OS (see Section 1.2.2.1) in this population. Fluoropyrimidine-based therapies (capecitabine, 5-FU) are the standard of care in mGC in general and were also the most frequent combination agents used in the ToGA trial (BO18255; see Section 1.2.2.1).

Furthermore, preclinical data suggest that the combination of trastuzumab emtansine and capecitabine has an additive effect (see Section 1.2.3).

A development program for trastuzumab emtansine is in place to seek approval for mGC indications. Capecitabine in combination with anti-HER2 agent is a proven efficacious regimen with a well-established safety profile in mGC. Trastuzumab emtansine and capecitabine might have overlapping toxicities and therefore a safety monitoring is in place to avoid exposing patients to harm. Therefore, exploring the benefit of combination therapy of trastuzumab emtansine and capecitabine in patients with mGC seems justified. Results from the Phase I part of the study in mGC will be used as supporting information for future studies in the indication.

# 2. <u>OBJECTIVES</u>

# 2.1 PHASE I: MTD FINDING OF TRASTUZUMAB EMTANSINE AND CAPECITABINE IN MBC

## 2.1.1 PRIMARY OBJECTIVE

 To determine the MTD of the combination of trastuzumab emtansine and capecitabine in patients with mBC

# 2.1.2 SECONDARY OBJECTIVES

- PK of trastuzumab emtansine and metabolites and capecitabine
- Safety of the combination of trastuzumab emtansine and capecitabine

ORR

# 2.2 RANDOMIZED PHASE II: EXPLORATION OF EFFICACY AND SAFETY IN MBC

### 2.2.1 PRIMARY OBJECTIVE

To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine in patients with mBC, as measured by ORR by RECIST v.1.1 per investigator local assessment

## 2.2.2 SECONDARY OBJECTIVES

Safety profile of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine

To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine in patients with mBC, as measured by:

- Time to response (TTR)
- DoR
- TTP
- Time to treatment failure (TTF)
- PFS
- CBR
- OS

# 2.3 PHASE I: MTD FINDING OF TRASTUZUMAB EMTANSINE AND CAPECITABINE IN MGC

#### 2.3.1 PRIMARY OBJECTIVE

To determine the MTD of the combination of trastuzumab emtansine and capecitabine in patients with mGC

# 2.3.2 SECONDARY OBJECTIVES

- PK of trastuzumab emtansine and metabolites and capecitabine
- Safety of the combination of trastuzumab emtansine and capecitabine
- ORR

# 3. STUDY DESIGN

# 3.1 DESCRIPTION OF STUDY

This is an international, multicenter Phase I/II dose finding study of two dosing schedules of trastuzumab emtansine and capecitabine combination therapy in HER2-positive mBC and locally advanced or patients with mGC.

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in a Phase I study in patients with mBC and locally advanced or mGC. The efficacy and safety of the combination in patients with mBC will also be explored in a randomized, open-label Phase II part of the study.

# 3.1.1 OVERVIEW OF STUDY DESIGN

# **Overview of Study Design**

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with HER2-positive mBC and locally advanced or mGC, using a Phase I design, followed by a randomized, openlabel Phase II part of the study to explore the efficacy and safety of the combination in patients with mBC. There will be no exploration of efficacy in the mGC cohort. Results from the Phase I in mGC will be used as supporting information for future studies in the indication.

Cohort 1 for patients with mBC will open first and MTD will be established. Once MTD is established, both randomized Phase II for patients with mBC and Cohort 2 for patients with mGC will open.

An overview of the study design is depicted in Figure 4.

# **Duration of Treatment and Patient Follow-up**

<u>Length of treatment:</u> All patients will be treated until disease progression, intolerable toxicity, withdrawal of consent, or death.

<u>Patient follow-up:</u> All patients will be followed-up until withdrawn consent, death, or up to a maximum of 2 years after the last patient was randomized in the Randomized Phase II part of the study, whichever occurs first.

# **Duration of Study, Database Closure and Data Reporting**

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to be 2 years for the Dose Finding and the Phase II/Exploration of Efficacy and Safety. The study will end after the follow-up period is completed, as defined above. Last patient last visit (LPLV) is defined as the last data collection point that can be either a clinic visit or a laboratory sample. At that time point, the database will be closed.

In the case that in Cohort 1 the Dose Level -2 is too toxic (> 1/6 of dose-limiting toxicity [DLT]), the combination may be considered unfeasible, recruitment will be closed and neither the Randomized Phase II nor mGC cohort will be opened. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the Steering Committee (SC).

Data may be reported at the end of each cohort i.e., once the MTD for Cohort 1 for mBC has been defined and the dose for Phase II/Exploration of Efficacy and Safety has been selected. The latest point to write the Clinical Study Report (CSR) will be 1 year after database closure.


If at the moment of study closure there are patients who have not progressed and are still receiving study treatment, they will be offered the possibility to continue treatment by enrolling in an extension study.

Figure 4 Overview of Study Design



<sup>&</sup>lt;sup>1</sup>Capecitabine doses are administered daily on Days 1 to 14 of the 3-week cycles

A schedule of assessments is provided in Appendix 1.

# 3.1.1.1 Overview of Phase I Design in Patients with mBC

An overview of the Phase I study design is depicted in Figure 5.

<sup>&</sup>lt;sup>2</sup>The MTD defined in mBC Phase I will be implemented in mBC Randomized Phase II and mGC Phase I

<sup>&</sup>lt;sup>3</sup> Cohort 2 will open to recruit patients with mGC once the MTD is defined in Phase I for patients with mBC. Dose Level 1 will not be explored in Cohort 2 (see also Section 3.3.2.1) mBC = metastatic breast cancer; mGC = metastatic gastric cancer; MTD = maximum tolerated dose; q3w = every 3 weeks; qw = weekly; T-DM1 = trastuzumab emtansine



Figure 5 Overview of Phase I Dose Finding Study Design

DLT = dose-limiting toxicity; MTD = maximum tolerated dose

# **Determination of the Maximum Tolerated Dose in Patients with mBC**

The trial will first investigate the feasibility of the combination of capecitabine and trastuzumab emtansine q3w in one cohort up to 18 patients, by deescalating the dose of capecitabine from 750 mg/m² bid to 650 mg/m² bid on Days 1 to 14 in cycles of 3 weeks with a 3 plus 3 classical Phase I design. Cohort 1 will open first and enroll patients with HER2-positive mBC.

# **Enrollment into Cohort 1**

# Dose finding in patients with mBC (Phase I)

According to the 3 plus 3 classical study design, Cohort 1 will start with the enrollment of 3 patients at Dose Level 1. Patients will be evaluated for DLTs as specified in DLT definition (see Section 5.1.3). The dose tested of trastuzumab emtansine will remain fixed at 3.6 mg/kg q3w and 3 dose levels of capecitabine administered bid on Days 1 to 14 in 3-week cycles will be tested.

The following doses will be explored in Cohort 1:

**Dose Level 1:** 750 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine

**Dose Level -1:** 700 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine


45

<sup>&</sup>lt;sup>1</sup> Repeat with the new dose level until the MTD is established

<sup>&</sup>lt;sup>2</sup> If Dose Level -2 is too toxic (> 1/6 DLT), the study will be terminated.
**Dose Level -2:** 650 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine

If Dose Level -2 is found to be too toxic (DLT > 1/6), the combination may be considered unfeasible, the recruitment will be closed and neither the Randomized Phase II nor mGC cohort will be opened. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the SC.

The following MTD determining rules will be applied during the Dose Finding treatment phase:

- Step 1: Three patients will be enrolled at Dose Level 1
- Step 2: The toxicity of Dose Level 1 will be monitored and the following actions taken:
  - a) If none of these 3 patients (0/3) experiences a DLT, the MTD will be established as the current dose level and will need to be confirmed in 3 more patients (to achieve ≤ 1/6 DLT at the current dose level)
  - b) If 1 of the initial 3 patients (1/3) experiences a DLT, additional 3 patients should be enrolled and treated at the same dose, i.e., Dose Level 1
  - c) If no more patients experience a DLT (1/6), the MTD will be established as the current dose level
  - d) If 1 or more patients experience a DLT (> 1/6), the dose will be deescalated to the next lower dose level. If no more than 1 patient experiences a DLT (≤ 1/6) after dose de-escalation, the dose will be considered the MTD and, following iDMC agreement, will be further explored in the Randomized Phase II part of the study. Dose re-escalation will not be allowed. If 2 or more patients experience DLT (> 1/6) after dose de-escalation, de-escalation should continue to the next lower dose level. Based on the DLT findings, the next dose level may be considered the MTD and, following iDMC agreement, be further explored in the Randomized Phase II part of the study or the study may be terminated if > 1/6 DLTs occur at Dose Level -2

In order to define the dose for the Randomized Phase II/Exploration of Efficacy and Safety part of the study, not only the DLTs during Cycle 1 will be evaluated but also all available safety information during the subsequent cycles. The dose level considered optimal will be the dose level selected to move forward with in the Phase II and mGC parts of the study.

Once the appropriate dose of study medication is established, the Randomized Phase II part of the study and Phase I, Cohort 2 will open as per Figure 4.

# 3.1.1.2 Overview of Phase II: Exploration of Efficacy and Safety in Patients with mBC

This part of the study will explore the efficacy and safety of the combination treatment of T-DM1 and capecitabine, at the established MTD, compared with T-DM1 alone in mBC patients.

Once the MTD has been defined to treat patients in Phase II, approximately 117 additional patients with mBC will be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to the Phase II part of the study; however, they will be followed-up until end of study (EOS).

Patients will be treated until disease progression/recurrence, intolerable toxicity, withdrawn consent, or death. If capecitabine needs to be discontinued for any reason, trastuzumab emtansine may continue, and the patient will be followed-up until EOS. In case of discontinuation of trastuzumab emtansine, patients will be followed-up until EOS.

All patients will be followed-up until withdrawn consent, death, or up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first.

See Section 3.1.1 for further information.

# 3.1.1.3 Overview of Phase I Design in mGC Patients

#### Determination of MTD in Patients with mGC

Cohort 2 will open when the capecitabine MTD is established for Cohort 1 and enroll patients with HER2-positive locally advanced and mGC. Trastuzumab emtansine will be administered qw at the fixed dose of 2.4 mg/kg and capecitabine will be started at the MTD defined for patients with mBC in Cohort 1. See Section 3.1.1 for further information.

#### **Enrollment into Cohort 2**

Cohort 2 will open with a 3 plus 3 classical design to investigate the feasibility of combination therapy of capecitabine and trastuzumab emtansine in Cohort 2 (enrolling up to 12 patients with mGC) by de-escalating the dose of capecitabine starting from the MTD determined in Cohort 1. In case the MTD was not established or the enrollment was stopped for Cohort 1, enrollment into Cohort 2 will not take place.

The dose levels for de-escalation of capecitabine will be the same as described for Cohort 1, except for Dose Level 1, which will not be explored in patients with mGC (see also Section 3.3.2.1).

If the MTD established in Cohort 1 is defined at Dose Level -1:

 This will be the starting dose in Cohort 2. If Dose Level -1 is well tolerated (DLT ≤ 1/6), this dose will be established as the MTD for mGC.  De-escalation: if Dose Level -1 is not tolerated in Cohort 2 (> 1/6 DLT), de-escalation will be to Dose Level -2.

If the MTD established in Cohort 1 is defined at Dose Level -2:

- This will be the starting dose in Cohort 2. If Dose Level -2 is well tolerated (DLT ≤ 1/6), this dose will be established as the MTD for mGC.
- De-escalation: if Dose Level -2 is not tolerated in Cohort 2 (> 1/6 DLT), the combination will be considered not feasible in mGC and Cohort 2 will be terminated. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on riskbenefit balance and agreement with the SC

#### 3.1.1.4 Number of Patients

Overall, it is anticipated that the maximum number of patients enrolled into the study will be approximately 147 patients.

### Phase I, Cohort 1: mBC

From a minimum of 6 to 18 patients will be enrolled into Cohort 1 to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with mBC.

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

For this part of the study, a total of approximately 117 patients with mBC will be randomized.

# Phase I, Cohort 2: mGC

After the MTD in Cohort 1 has been established, 3–12 patients will be enrolled into Cohort 2 to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with mGC.

#### 3.1.1.5 Number of Centers

This is a multicenter, international study.

#### 3.1.2 STEERING COMMITTEE

A SC has been established for this study. Initially, it is composed of the investigators participating in the Phase I, Cohort 1 part of the study and one medical representative and one statistician of the Sponsor. The study design and DLT has been developed by the SC. See SC Charter for further information.

The SC will collectively review the status of the ongoing patients on a regular basis. The SC will also review in due course all available efficacy data and PK information to ensure that safety information is in the context of risk-benefit and that dosing is also related to exposure to the drug.

The SC will adjudicate in cases of DLTs that are not covered by the existing DLT criteria.

#### 3.1.3 INDEPENDENT DATA MONITORING COMMITTEE

An independent data monitoring committee (IDMC) will be established for the Randomized Phase II part of the study. The IDMC will review the safety outcomes for patients enrolled in Phase I, Cohort 1 and advise whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 20 and 60 patients have received at least 3 cycles (Cycle 3 Day 1) of treatment in the Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II of the study or as requested.

#### 3.2 END OF STUDY

End of study (EOS) is defined as LPLV at the end of the follow-up period, as defined in Section 3.1.1. This will be the last data collection point, which can be a clinic visit or a laboratory sample. LPLV is expected to occur approximately 2 years after the last patient has been enrolled into the trial.

# 3.3 RATIONALE FOR STUDY DESIGN

# 3.3.1 RATIONALE FOR PATIENT GROUP SELECTION

Nonclinical studies indicate that the sensitivity of cancer cells to trastuzumab emtansine requires HER2 overexpression, and measurement of such expression is a standard of care in determining eligibility for trastuzumab therapy (see the Herceptin® national prescribing information). Measurement of HER2 gene amplification has traditionally been performed using IHC measurement. HER2 gene amplification determined by FISH has also proven to be a reliable method for demonstrating HER2-positive status (Press et al. 2005).

This study will enroll patients diagnosed with the disease, to which the combination is intended. The combination of anti-HER2 agent and capecitabine has shown to be efficacious in both mBC (von Minckwitz et al. 2011; Geyer et al. 2006) and mGC (Bang et al. 2010), and capecitabine is a standard of care treatment for both diseases. Both diseases have been shown to benefit from anti-HER2 treatment; therefore, all patients must be diagnosed with HER2-positive disease. Patients with incurable mBC and locally advanced or mGC, whose tumors are positive for HER2 overexpression, represent the patient population eligible for study enrollment.

#### 3.3.1.1 Rationale for Phase I

The study design of 3 plus 3 Phase I is a well-established and well-known method for Phase I studies. PK parameters will be collected and analyzed in order to investigate the PK interaction of the drugs under investigation. Since both agents are administered at efficacious doses, the risk of enrolling patients at the sub-optimal doses is minimal.

Following review of preliminary data from Cohort 1 of this study by the SC for patients enrolled to receive 750 mg/m² capecitabine, where 2 DLTs were observed in 6 evaluable patients, it was decided not to explore dose levels of capecitabine higher than 750 mg/m². According to the investigator assessment and the SC recommendation, the available evidence shows an acceptable positive risk-benefit in all 7 patients treated at Dose Level 1.

As of 7 August 2013, five patients remain on treatment, with a follow-up period of 4 to 8 months. Of the two patients who have discontinued treatment, one patient's disease has progressed, and the other discontinuation was based on the investigator's decision, following the central confirmation, that the patient's disease was HER2-negative. Considering the available safety data for all patients (maximum number of cycles is 12), the combination of capecitabine and T-DM1 is well tolerated, except for increases in transaminases and hand-foot syndrome. Dose modifications of T-DM1 and/or capecitabine have allowed those patients to continue on treatment. Of note, no SAE has been reported in 6 patients. Latest tumor response data show 2 patients with PR and 4 patients with SD. Any required dose modifications (dose reductions) are allowed for each individual drug as described in Sections 5.1.5.1 and 5.1.5.2 and are in line with the trastuzumab emtansine Investigator's Brochure and Xeloda® Summary of Product Characteristics.

The combination of T-DM1 and capecitabine will be evaluated with a deescalation study design. Patients who are currently receiving the combination of T-DM1 and capecitabine 750 mg/m² can continue to receive the dose as per protocol until there is no longer evidence of positive risk-benefit as per investigator assessment and SC endorsement.

#### 3.3.1.2 Rationale for Randomized Phase II

Randomized Phase II part of the study is designed to provide an estimation of the treatment effect of the combination, at the selected MTD, compared with T-DM1 alone.

The patient data will be stratified by previous anti-cancer treatment (excluding single-agent hormones) for the treatment of metastatic disease (1 or >1 prior lines of treatment). The stratified data will be compared with data from historical studies of single-agent trastuzumab emtansine in similar patient populations. This will allow a more robust evaluation of the added treatment effect of Xeloda® within the combination treatment.

A 2:1 randomization will be applied to allow more patients being exposed to the combination of T-DM1 and capecitabine. This will enable a more thorough assessment of the corresponding safety profile.

In addition, it will provide important information on the longer-term safety of the combination.

# 3.3.2 RATIONALE FOR INVESTIGATIONAL MEDICINAL DOSE SELECTION

#### 3.3.2.1 In Patients with mBC

In study TDM3569g, the MTD of trastuzumab emtansine administered by IV infusion q3w was 3.6 mg/kg. As described in Section 1.2, clinical activity has been observed at a dose of 3.6 mg/kg q3w in two Phase II studies of single-agent trastuzumab emtansine in patients with advanced heavily pre-treated HER2-positive mBC (protocol TDM4258g and protocol TDM4374g) and in patients who had not received prior chemotherapy for metastatic disease (TDM4450g).

Capecitabine doses have been selected as being in the range of efficacious doses for single-agent or combination use. The doses selected are within the dosing range included in the Xeloda<sup>®</sup> Summary of Product Characteristics (SmPC) and therefore are considered to be efficacious.

#### 3.3.2.2 In Patients with mGC

In the ToGA study (BO18255: trastuzumab in combination with chemotherapy in mGC), patients with higher drug exposure had a greater benefit compared with those with lower exposure (Yang et al. 2011). As a consequence, a randomized, open-label, multicenter Phase IIIb study comparing two trastuzumab dosing regimens, each in combination with cisplatin/capecitabine chemotherapy, as first-line therapy in patients with HER2-positive metastatic gastric or GEJ adenocarcinoma is being conducted (Study BO27798).

In TDM3569g (see Section 1.2.1.1), the qw administration of 2.4 mg/kg of trastuzumab emtansine resulted in higher exposure (see Section 1.2.1.7) (Krop et al. 2008). Therefore, this dose may result in larger clinical benefit for patients with mGC. Trastuzumab emtansine at 2.4 mg/kg qw is being tested in the BO27952 study.

In Cohort 2, the starting dose of capecitabine will be the MTD from Cohort 1 (mBC) in order to minimize the exposure of patients to sub-optimal treatment. The dose of capecitabine can be de-escalated if needed.

#### 3.3.2.3 Rationale for Duration of Treatment

Treatment will be given until disease progression or unacceptable toxicity (see Section 3.1.1 for full information). As of 1 January 2010, of 237 patients enrolled in studies TDM3569g, TDM4258g, and TDM4374g receiving trastuzumab emtansine at 3.6 mg/kg, approximately 30% have tolerated more than 12 cycles, with 14.8% having received more than 17 cycles. Twenty patients (8.4%) have discontinued trastuzumab emtansine due to AEs and 24 patients (10.1%) required dose reductions in trastuzumab emtansine because of AEs. In the absence of intolerable toxicity, patients with mBC are generally treated until disease progression.

Capecitabine will be given until disease progression, as per Xeloda<sup>®</sup> national prescribing information.

# 3.3.3 PHARMACOKINETIC SAMPLING RATIONALE

The PK sampling rationale is to characterize the PK of trastuzumab emtansine, total trastuzumab, and DM1, to assess potential drug-drug interaction when trastuzumab emtansine is given in combination with capecitabine, and to explore potential correlations between drug exposure and measures of both efficacy (ORR) and toxicity (alanine transaminase [ALT]/AST, platelets, etc.), if data allow.

### 3.4 OUTCOME MEASURES

# 3.4.1 PHASE I: MBC

# 3.4.1.1 Primary Efficacy Outcome Measure

The main objective for Phase I is to determine the MTD of capecitabine when combined with trastuzumab emtansine.

# 3.4.1.2 Secondary Efficacy Outcome Measure

The secondary outcome is ORR, based on best overall response (BOR) rate as per RECIST v.1.1; per investigator local assessment.

# 3.4.1.3 Primary Safety Outcome Measure

The primary safety outcome measure is to establish the MTD. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination and will be summarized for each treatment dosage.

# 3.4.1.4 Secondary Safety Outcome Measures

Safety endpoints will be summarized for each treatment dosage:

- Incidence, nature, and severity of AEs, as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v. 4.0
- Incidence, nature, and severity of SAEs, as per NCI CTCAE v. 4.0
- Incidence and nature of AEs equal or higher than Grade 3
- Incidence, nature, and severity of AEs of special interest (AESIs), as per NCI CTCAE v. 4.0
- Premature withdrawal from study medication
- Abnormal laboratory values
- LVEF
- Exposure to study medication
- Concomitant medications and physical examination

#### 3.4.1.5 Pharmacokinetic Outcome Measures

The PK outcome measures to be assessed in patients receiving trastuzumab emtansine and capecitabine will include:

- Serum concentrations of trastuzumab emtansine (conjugated drug) and total trastuzumab (free and conjugated to DM1)
- Plasma concentration of DM1
- Plasma concentration of capecitabine and its active metabolite 5-FU

# 3.4.2 RANDOMIZED PHASE II: EXPLORATION OF EFFICACY AND SAFETY IN MBC

The primary and secondary efficacy outcome measures will be presented for each treatment group.

# 3.4.2.1 Primary Efficacy Outcome Measure

The primary outcome measure is ORR by investigator assessment, based on BOR (defined as the best response recorded from the start or randomization into Phase II part of the study and until disease progression or recurrence, death, withdrawal of consent, or EOS, whichever occurs first) as per RECIST v.1.1 provided in Appendix 3.

# 3.4.2.2 Secondary Efficacy Outcome Measures

Secondary outcomes include:

- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

# 3.4.2.3 Primary Safety Outcome Measure

A primary safety outcome is defined only for Phase I, and will be presented for both treatment groups.

# 3.4.2.4 Secondary Safety Outcome Measures

Again, the summary of safety endpoints will be presented for each treatment group:

- Incidence, nature, and severity of AEs, as per NCI CTCAE v. 4.0
- Incidence, nature, and severity of SAEs, as per NCI CTCAE v. 4.0
- Incidence and nature of AEs equal or higher than Grade 3
- Incidence, nature, and severity of AESIs, as per NCI CTCAE v. 4.0
- Premature withdrawal from study medication
- Abnormal laboratory values
- LVEF

- Exposure to study medication
- Concomitant medications and physical examination

#### 3.4.2.5 Pharmacokinetic Outcome Measures

Not applicable for Phase II.

#### 3.4.3 Phase I: MGC

# 3.4.3.1 Primary Efficacy Outcome Measure

The main objective for Phase I is to determine the MTD of capecitabine when combined with trastuzumab emtansine.

# 3.4.3.2 Secondary Efficacy Outcome Measure

The secondary outcome is ORR, based on BOR rate as per RECIST v.1.1; based on investigator assessment.

# 3.4.3.3 Primary Safety Outcome Measure

The primary outcome measure is to establish MTD. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination and will be summarized for each treatment dosage.

# 3.4.3.4 Secondary Safety Outcome Measures

Safety endpoints will be summarized for both treatment phases: Dose Finding and Exploration of Efficacy. Again, the summary of safety endpoints will be presented for each treatment dosage:

- Incidence, nature, and severity of AEs, as per NCI CTCAE v. 4.0
- Incidence, nature, and severity of SAEs, as per NCI CTCAE v. 4.0
- Incidence and nature of AEs equal or higher than Grade 3
- Incidence, nature, and severity of AESIs, as per NCI CTCAE v. 4.0
- Fatal cases and causes of death
- Laboratory parameters
- LVEF
- Treatment exposure

#### 3.4.3.5 Pharmacokinetic Outcome Measures

The PK outcome measures to be assessed in patients receiving trastuzumab emtansine and capecitabine will include:

- Serum concentrations of trastuzumab emtansine (conjugated drug) and total trastuzumab (free and conjugated to DM1)
- Plasma concentration of DM1
- Plasma concentration of capecitabine and its active metabolite 5-FU

# 4. MATERIALS AND METHODS

# 4.1 PATIENTS

#### 4.1.1 PATIENTS WITH MBC

This study will enroll patients with HER2-positive BC with histologically or cytologically confirmed metastatic disease, which are amenable for combination treatment with trastuzumab emtansine and capecitabine.

Patients with mBC must have received at least one treatment regimen, which includes a chemotherapy and trastuzumab agent. Only patients whose HER2 tumor status was locally scored as IHC 3+ or ISH positive will be permitted for both study parts (Phase I and II).

# 4.1.2 MGC PATIENTS

This study will enroll patients with HER2-positive GC with histologically or cytologically confirmed inoperable locally advanced or metastatic disease, which are amendable for combination treatment with trastuzumab emtansine and capecitabine.

Patients with mGC must have not received prior chemotherapy for advanced/metastatic disease, and only patients with HER2-positive primary tumor or metastasis as assessed by central laboratory will be allowed to enroll in the Dose Finding part for this disease in this study.

#### 4.1.3 INCLUSION CRITERIA

# 4.1.3.1 For Patients with mBC

Patients must meet the following criteria for study entry:

- 1. Age ≥ 18 years old
- 2. Signed informed consent prior to any study specific procedure
- 3. Able and willing to comply with protocol
- 4. Negative serum pregnancy test for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential.
- 5. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 6 months after the last dose of study treatment (see Section 5.2.4).
- 6. ECOG performance status of 0, 1, or 2

#### 7. Blood:

- a) Platelet count > 100,000 cells/mm<sup>3</sup>
- b) International normalized ratio (INR) < 1.5
- c) Absolute neutrophil count (ANC) > 1,500 cells/mm<sup>3</sup>
- d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.

#### 8. Liver function:

- a) Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
- b) Serum glutamic oxaloacetic transaminase (SGOT)/AST and serum glutamic pyruvic transaminase (SGPT)/ALT ≤ 2.5 × the ULN
- c) Alkaline phosphatase ≤ 2.5 × the ULN. Patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × the ULN
- d) Evidence of stable liver function during the month prior to enrollment with liver function tests' (LFTs) fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN

#### 9. Renal function:

a) Serum creatinine of < 177 μmol/L or calculated creatinine CL > 50 mL/min. I urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate ≤ 1 g of protein/24 hours

#### 10. Cardiac function:

- a) LVEF ≥ 50% by echocardiogram (ECHO) or multiple-gated acquisition (scan) (MUGA)
- 11. Histologically or cytologically confirmed BC
- 12. HER2-positive disease IHC 3+ or ISH positive
- 13. Tumor block or 15 slides available for retrospective central confirmation of HER2-positivity (central confirmation not necessary for enrollment).
- 14. mBC with at least one measurable lesion according to RECIST v.1.1
- 15. Disease progression on at least one regimen containing trastuzumab and chemotherapy
- 16. Patients must have recovered from previous treatments

# 4.1.3.2 For Patients with mGC

Patients must meet the following criteria for study entry:

- 1. Age ≥ 18 years old
- 2. Signed informed consent prior to any study specific procedure
- 3. Able and willing to comply with protocol
- Negative serum pregnancy test for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of


- amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential
- 5. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 6 months after the last dose of study treatment (see Section 5.2.4)
- 6. ECOG performance status of 0, 1, or 2
- 7. Blood:
  - a) Platelet count > 100,000 cells/mm3
  - b) INR < 1.5
  - c) ANC  $> 1,500 \text{ cells/mm}^3$
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 8. Liver function:
  - a) Total bilirubin ≤ 1.5 × ULN
  - b) SGOT/AST and serum glutamic pyruvic transaminase (SGPT)/ALT ≤ 2.5 × the ULN
  - c) Alkaline phosphatase ≤ 2.5 × the ULN. Patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × the ULN
  - d) Evidence of stable liver function in the month prior to enrollment with LFTs fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN
- 9. Renal function:
  - a) Serum creatinine of < 177 μmol/L or calculated creatinine CL > 50 mL/min. I urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate ≤ 1 g of protein/24 hours
- 10. Cardiac function:
  - a) LVEF ≥ 50% by ECHO or MUGA
- 11. Histologically or cytologically confirmed mGC or locally advanced GC
- 12. HER2-positive tumor (primary tumor or metastatic lesion), defined as either IHC 3+ alone or IHC 2+ in combination with ISH+, prospectively confirmed by a Sponsor-designated central laboratory prior to enrollment. ISH positivity is defined as a ratio of ≥ 2.0 for the number of HER2 gene copies to the number of signals for CEP17.
  - a) Archival tumor samples obtained from primary or metastatic sites are acceptable.

- b) Invasive tumor for central confirmation of HER2 status is required.
- c) A formalin-fixed paraffin-embedded (FFPE) tissue block with at least 5 mm of invasive tumor for central confirmation is preferred.

If FFPE tissue blocks (or partial block) are unavailable due to country or site regulations, a minimum of 8 freshly cut unstained slides MUST be available for central review of HER2 status.

13. Inoperable locally advanced or mGC

#### 4.1.4 EXCLUSION CRITERIA

#### 4.1.4.1 For Patients with mBC

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half-lives, whatever is longest
  - b) Hormonal therapy within 14 days
  - c) Trastuzumab within 21 days
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received prior trastuzumab emtansine
- 3. Prior treatment with capecitabine
- 4. History of severe and unexpected reactions to fluoropyrimidine or with known hypersensitivity to fluorouracil
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogues, such as brivudine
  - b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>
  - b) Epirubicin > 900 mg/m<sup>2</sup>
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 28 days of first study drug administration
- 9. Current peripheral neuropathy of Grade ≥ 3 per the NCI CTCAE, v. 4.0

10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above

- 11. Current unstable ventricular arrhythmia requiring treatment
- 12. History of symptomatic CHF (New York Heart Association [NYHA] Classes II-IV)
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
- 15. Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation
- 20. Current known active infection with human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C virus (HBV/HCV)
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Lapatinib ≤ 14 days before first study drug administration
- 22. Previous radiotherapy for the treatment of unresectable, locally advanced/recurrent or mBC is not allowed if:
  - a) The last fraction of radiotherapy has been administered within 14 days prior to first study drug administration.
  - b) More than 25% of marrow-bearing bone has been irradiated.
  - c) The patient has not recovered from any resulting acute toxicity to Grade ≤ 1 prior to first study drug administration.
- 23. No signs and symptoms suggestive that the patient has dihydropyrimidine dehydrogenase (DPD) deficiency

#### 4.1.4.2 For Patients with mGC

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half-lives, whatever is longest
  - b) Hormonal therapy within 14 days

242

- c) Trastuzumab within 21 days
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received prior trastuzumab emtansine
- 3. Prior treatment with capecitabine
- 4. History of severe and unexpected reactions to fluoropyrimidine or with known hypersensitivity to fluorouracil
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogues, such as brivudine
  - b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>
  - b) Epirubicin > 900 mg/m<sup>2</sup>
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m<sup>2</sup> doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 28 days of first study drug administration
- 9. Current peripheral neuropathy of Grade ≥ 3 per the NCI CTCAE, v. 4.0
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above
- 11. Current unstable ventricular arrhythmia requiring treatment
- 12. History of symptomatic CHF (NYHA Classes II-IV)
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
- 15. Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)

- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation
- 20. Current known active infection with HIV, HBV, and/or HCV
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Previous chemotherapy for advanced/metastatic disease
  - a) Prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrollment into the study
- 22. No signs and symptoms suggestive that the patient has DPD deficiency
- 23. Lapatinib ≤ 14 days before first study drug administration

# 4.1.5 PATIENT REPLACEMENT POLICY

None of the patients in the Phase I part of the study may be replaced unless approved by the entire SC.

# 4.2 METHOD OF TREATMENT ASSIGNMENT

In the Randomized Phase II part of the study, patients will be randomized to receive either the combination of T-DM1 and capecitabine or T-DM1 alone. The 2:1 randomization ratio will be applied to allow more patients being exposed to the combination treatment and to enable a more thorough assessment of the corresponding safety profile.

This is an open-label study; therefore, no blinding will be used.

# 4.3 STUDY TREATMENT

# 4.3.1 FORMULATION, PACKAGING, AND HANDLING

#### 4.3.1.1 Trastuzumab Emtansine

Trastuzumab emtansine is provided as a single-use, lyophilized formulation in a colorless 20 mL Type I glass vial containing 160 mg of trastuzumab emtansine, closed by means of a FluroTec coated stopper and an overseal with flip-off cap. Upon receipt of trastuzumab emtansine, vials should be refrigerated at 2–8°C (36–46°F) until use. THE VIAL MUST NOT BE FROZEN OR SHAKEN. Trastuzumab emtansine must be stored in the original carton to protect it from light. Do not use the product beyond the expiration date provided by the manufacturer. The reconstituted product contains no preservative and is intended for single use only. Any remaining medication should be discarded.

All vials of trastuzumab emtansine should be handled by appropriately trained site staff wearing gloves and using appropriate procedures in place at the

clinical site for preparation of chemotherapeutic drugs. Vials should be visually inspected upon receipt to ensure that they are intact without exterior contamination. Discard any cracked vials and report vials with surface contamination to the clinical site manager for assessment.

The lyophilized product should be reconstituted using sterile water for injection (SWFI). Using a new syringe, 8 mL SWFI should be added to the vial and the vial swirled gently until the product is completely dissolved. The vial should not be shaken. The resulting product contains 20 mg/mL trastuzumab emtansine, 10 mM sodium succinate, pH 5.0, 60 mg/mL sucrose, and 0.02% (w/v) polysorbate 20. Each 20 mL vial contains enough trastuzumab emtansine to allow delivery of 160 mg trastuzumab emtansine. The reconstituted product contains no preservative and is intended for single use only.

The vial should be inspected to ensure the reconstituted product is a clear colorless solution, and is free of particulates before proceeding. Drug from any vial that appears abnormal upon inspection should not be administered to patients. Using a new syringe, the indicated volume of trastuzumab emtansine solution should be removed from the vial(s) and added to the IV bag containing at least 250 mL of 0.45% sodium chloride (preferred) or 0.9% sodium chloride injection and gently inverted to mix the solution. A 0.22 micron non-protein adsorptive polyethersulfone in line filter is recommended when using 0.45% sodium chloride and required when using 0.9% sodium chloride injection. The solution of trastuzumab emtansine should not be shaken.

The solution of trastuzumab emtansine for infusion should be used immediately. If not used immediately, storage times should not be longer than 24 hours at 2–8°C (36–46°F) for solutions of trastuzumab emtansine diluted in polyvinyl chloride (PVC) or latex free PVC-free polyolefin, polypropylene, or polyethylene bags containing 0.45% or 0.9% Sodium Chloride for Injection.

For additional details, please refer to the current version of the trastuzumab emtansine Investigator's Brochure.

# 4.3.1.2 Capecitabine

The following information has been obtained from the Xeloda<sup>®</sup> EU SmPC and U.S. Xeloda<sup>®</sup> Package Insert.

Capecitabine is available as biconvex, oblong, film-coated tablets, available as follows:

- 150 mg tablets: color, light peach; engraving, XELODA on one side, 150 on the other; packs of 60
- 500 mg tablets: color, peach; engraving, XELODA on one side, 500 on the other; packs of 120

Capecitabine tablets should not be stored above 30°C.

# 4.3.2 DOSAGE AND ADMINISTRATION

#### 4.3.2.1 For Patients with mBC

#### **Trastuzumab Emtansine**

Trastuzumab emtansine will be administered on Day 1 of a 3-week cycle q3w at a dose of 3.6 mg/kg IV (see Appendix 1). The total dose will be calculated based on the patient's weight on Day 1 (or up to 3 days before) of each cycle with no upper limit.

If the timing of trastuzumab emtansine coincides with a holiday that precludes the procedure, the procedure should be performed within 3 business days of the scheduled date and, when possible, on the earliest following date, with subsequent protocol-specified procedures rescheduled accordingly.

The first infusion of trastuzumab emtansine will be administered over 90 minutes (±10 minutes). Infusions may be slowed or interrupted for patients experiencing infusion-associated symptoms. Vital signs must be assessed before and after dose administration. Following the initial dose, patients will be observed for at least 90 minutes for fever, chills, or other infusion-associated symptoms. If prior infusions were well tolerated (without any signs or symptoms of infusion reactions), subsequent doses of trastuzumab emtansine may be administered over 30 minutes (±10 minutes), with a minimum 30-minute observation period following infusion. Local health authority guidelines must be followed with regard to further observation and monitoring, if applicable.

Pre-medication for nausea and infusion reactions (e.g., acetaminophen or other analgesics, antihistamines such as diphenhydramine, or corticosteroids) may be given at the investigator's discretion.

# Capecitabine

Capecitabine will be administered twice a day, orally for 14 days followed by a 7-day rest period at the Dose Levels 1 to -2 described in the "Study Design" Section 3.1.1. Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Capecitabine doses can be delayed for up to 4 hours, while keeping the minimal interval of 8 hours between the doses.

Rounding of the dose, based on 150 and 500 mg strength tablets, will be allowed to the nearest dose per patient body surface area (BSA).

If a dose is missed, the patient should skip that dose. The patient should not double the dose during the next administration.

Guidelines for dosage modification and treatment interruption or discontinuation are provided in Section 5.1. For this part of the study, the MTD established in Phase I, Cohort 1 will be used as a starting dose.

#### 4.3.2.2 For Patients with mGC

#### **Trastuzumab Emtansine**

Trastuzumab emtansine will be administered on Day 1 of a qw cycle qw at a dose of 2.4 mg/kg IV (see Appendix 1). The total dose will be calculated based on the patients weight on Day 1 (or up to 3 days before) of each cycle with no upper limit.

Administration time and observation period will be performed as described in Section 4.3.2.1 for trastuzumab emtansine.

Guidelines regarding timing delays and infusion times are the same as for patients with mBC, as is the accepted pre-medication.

# Capecitabine

Capecitabine will be administered twice a day, orally, for 14 days followed by a 7-day rest period at the dose level that was determined during the Dose Finding part of the study in patients with mBC as the MTD in Cohort 1. Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Capecitabine doses can be delayed for up to 4 hours, while keeping the minimal interval of 8 hours between the doses.

If a dose is missed, the patient should skip that dose. The patient should not double the dose the next administration.

Guidelines for dosage modification and treatment interruption or discontinuation are provided in Section 5.1.

#### 4.3.3 INVESTIGATIONAL MEDICINAL PRODUCT ACCOUNTABILITY

All investigational medicinal products (IMPs) required for completion of this study (trastuzumab emtansine and capecitabine) will be provided by the Sponsor. The investigational site will acknowledge receipt of IMPs, using the interactive voice/web recognition system (IxRS) to confirm the shipment condition and content. Any damaged shipments will be replaced.

IMPs will either be disposed of at the study site according to the study site's institutional standard operating procedure or returned to the Sponsor with the appropriate documentation. The site's method of IMP destruction must be agreed upon by the Sponsor. The site must obtain written authorization from the Sponsor before any IMP is destroyed, and IMP destruction must be documented on the appropriate form.

Accurate records of all IMPs received at, dispensed from, returned to, and disposed of by the study site should be recorded on the Drug Inventory Log.

#### 4.3.4 POST-TRIAL ACCESS TO EXTENSION STUDY

Post-trial access of trastuzumab emtansine and capecitabine will be performed as described in Section 3.1.1, *Treatment of Patients and Database Closure*. In case a patient decides to withdraw from the study, no post-trial access will be granted. Currently, the Sponsor does not have any plans to

Study MO28230

provide other study interventions to patients after conclusion of the study or any earlier patient withdrawal.

# 4.4 CONCOMITANT AND EXCLUDED THERAPIES

#### 4.4.1 PERMITTED THERAPY

Concomitant therapy and pre-medication are defined as non-IMPs.

Concomitant therapy includes any prescription medication, over-the-counter preparation, or herbal therapy between the 14 days preceding first treatment and the Study Treatment Discontinuation Visit. Afterwards, only anti-cancer therapies will be collected as part of the survival follow-up period.

Pre-medication is allowed according to standard practice guidelines.

No pre-medication for the first infusion of trastuzumab emtansine is required; however, pre-medication is allowed at the investigator's discretion.

Concomitant use of erythropoiesis stimulating agents is allowed if clinically indicated in accordance with local prescribing guidelines.

Palliative radiotherapy may be permitted to treat pre-existing painful bone metastases or to treat brain metastases (for patients who have disease control outside of the brain). Please contact the Medical Monitor for approval. If the Medical Monitor cannot be reached because of time zone differences, radiotherapy may be administered, but the Medical Monitor should still be informed.

Other medications considered necessary for the patient's safety and well being may be given at the discretion of the investigator. Use of bisphosphonates or denosumab is permitted for the control of bone pain, prevention and/or treatment of bony metastases, and treatment of osteoporosis. If bisphosphonates are required for the treatment of symptomatic malignancy-associated hypercalcemia, tumor assessments should be performed to assess for potential disease progression.

#### 4.4.2 PROHIBITED THERAPY

Use of the therapies described below is prohibited during the study prior to discontinuation of study treatment (collectively, these will be referred to as non-protocol therapy).

Any therapies intended for the treatment of cancer, other than trastuzumab emtansine, whether they are approved by national health authorities or experimental, including cytotoxic chemotherapy, immunotherapy, hormonal therapy (other than megestrol acetate), and biologic or targeted agents (other than granulocyte colony-stimulating factor and erythropoiesis stimulating agents), are prohibited.

Radiotherapy for unequivocal disease progression is not permitted while on study treatment, with the exception of new brain metastases or isolated progression of previously treated brain lesions. Patients who have disease control outside of the brain, defined as continued PR or CR of any duration, or SD for  $\geq 3$  months, but who have developed brain metastases that are treatable with radiation will be allowed to continue to receive study therapy until they either experience systemic progression of their disease and/or further progression in the brain that cannot be treated with additional radiation. Patients must not miss more than one cycle of study treatment for the treatment of their brain metastases and must have an ECOG performance status of 0, 1, or 2 to continue on therapy. The Medical Monitor should be informed before a decision is made to resume study treatment after radiotherapy for brain metastases.

# 4.5 STUDY ASSESSMENTS

All patients will be closely monitored for safety and tolerability during all cycles of therapy and at the safety follow-up visit:

- Visits will be based on a q3w cycle for mBC
- Visits will be based on a qw cycle for mGC

Study assessments are outlined in this section and in Appendix 1.

# 4.5.1 DESCRIPTION OF STUDY ASSESSMENTS

All patients will be closely monitored for safety and tolerability during all cycles of therapy and at the Study Treatment Discontinuation Visit. Patients should be assessed for toxicity prior to each dose; dosing will occur only if the clinical assessment and local laboratory test values are acceptable. Trastuzumab emtansine will be administered either in q3w cycles (patients with mBC) or qw cycles (patients with mGC) if no additional time is required for reversal of toxicity. Dose delays and dose reductions will be allowed for trastuzumab emtansine as outlined in Section 5.1.5.

If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend that precludes the procedure within the allotted window, the procedure should be performed on the nearest following date (i.e., within 3 business days).

# 4.5.1.1 Medical History and Demographic Data

Medical history includes clinically significant diseases, surgeries, cancer history (including prior cancer therapies and procedures), smoking history, use of alcohol and drugs of abuse, and all medications (e.g., prescription drugs, over-the-counter drugs, herbal/homeopathic remedies, nutritional supplements) used by the patient within 14 days prior to the screening visit.

Demographic data will include age, sex, and self-reported race/ethnicity.

# 4.5.1.2 Vital Signs

Vital signs will include measurements of weight, respiratory rate, heart rate, blood pressure, and temperature. Abnormal or significant changes to vital signs from baseline should be recorded as AEs, if appropriate.

# 4.5.1.3 Physical Examinations

A complete physical examination should include the evaluation of head, eye, ear, nose, and throat; cardiovascular; dermatological; musculoskeletal; respiratory; gastrointestinal; and neurological systems. Changes from baseline abnormalities should be recorded at each subsequent physical examination. New or worsened abnormalities should be recorded as AEs if appropriate.

As part of tumor assessment, physical examinations should also include the evaluation of the presence and degree of enlarged lymph nodes, hepatomegaly, and splenomegaly.

Limited physical examinations will be symptom-directed.

# 4.5.1.4 Tumor and Response Evaluations

Measurable and unmeasurable disease must be documented at screening and re-assessed at each subsequent tumor evaluation. Tumor assessments with computed tomography (CT) or magnetic resonance imaging (MRI) scans of the chest, abdomen, and pelvis are to be performed as described in Appendix 1, Schedule of Assessment. CT or MRI of the brain and baseline radioisotope bone scan must be obtained at screening. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to first treatment the bone scan does not need to be repeated and non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Tumor assessments should include an evaluation of all known and/or suspected sites of disease, whenever possible. Patients should have lesions selected that can be evaluated at every tumor assessment. The same radiographic procedure used at screening must be used throughout the study (e.g., the same contrast protocol for CT scans). Response assessments will be assessed by the investigator, based on physical examinations, CT or MRI scans, and bone scans using RECIST v. 1.1 (see Appendix 3). In the event a positron emission tomography (PET)/CT scanner is used for tumor assessments, the CT portion of the PET/CT must meet criteria for diagnostic quality. For patients who continue study treatment after isolated brain progression, the frequency of follow-up scans is at the discretion of the investigator.

At the investigator's discretion, CT scans, MRI scans, and/or bone scans may be obtained at any time when clinically indicated or if PD is suspected. If a bone scan cannot be performed during the course of the study because of the unavailability of the Tc-99m isotope, the investigator may choose an alternative imaging modality (see Appendix 4).

Radiographic imaging should always be performed rather than clinical examination unless the lesion(s) being followed cannot be imaged but are assessable by clinical examination. In applying RECIST, documentation by color photography including a ruler to estimate the size of the lesion is recommended.

# 4.5.1.5 Laboratory Assessments

#### For Patients with mBC:

# **Local Laboratory Assessments:**

- Hematology, biochemistry, coagulation, urinalysis, and pregnancy testing
- Prospective or retrospective HER2 status. Patients will be enrolled based on local results.

# **Central Laboratory Assessments:**

- Retrospective HER2 status. Retrospective central confirmation will not impact the treatment decisions or primary endpoint of Phase I, Cohort 1 and will be used to validate efficacy analyses in Phase I and to censor the efficacy population for the Randomized Phase II part of the study
- PK assays:
- Serum trastuzumab emtansine concentration and total trastuzumab using a validated immunoassay
- Serum capecitabine and 5-FU PK samples
- Plasma concentration of DM1 using a validated liquid chromatography electrospray tandem mass spectrometry (LC-MS/MS) method

#### For Patients with mGC:

#### **Local Laboratory Assessments:**

Hematology, biochemistry, coagulation, urinalysis, and pregnancy testing

### **Central Laboratory Assessments:**

- Prospective HER2 status. Patients will be enrolled based on the central testing results
- PK assays:
- Serum trastuzumab emtansine concentration and total trastuzumab using a validated immunoassay
- Serum capecitabine and 5-FU PK samples
- Plasma concentration of DM1 using a validated liquid chromatography electrospray tandem mass spectrometry (LC-MS/MS) method

#### 4.5.1.6 Electrocardiograms

A 12-lead ECG should be obtained at baseline and be printed and kept with the patient's record.

#### 4.5.1.7 ECOG Performance Status

Performance status will be measured using the ECOG performance status scale (see Appendix 6).

It is recommended, where possible, that a patient's performance status be assessed by the same person throughout the study.

Performance status will be assessed according to the schedule of assessments (see Appendix 1)

#### 4.5.1.8 ECHO/MUGA

ECHO is the preferred modality because of the global technetium (Tc-99m) shortage (see Appendix 4). The same method used at screening should be used throughout the study.

#### 4.5.2 TIMING OF STUDY ASSESSMENTS

# 4.5.2.1 Screening and Pretreatment Assessments

Written informed consent for participation in the study must be obtained before performing any study specific screening tests or evaluations. Informed Consent Forms for enrolled patients and for patients who are not subsequently enrolled will be maintained at the study site.

Once the patient has signed the Informed Consent Form, the investigator (or his designee) will call the IxRS to obtain the screening number for the patient prior to Cycle 1, Day 1.

Results of standard of care tests or examinations performed prior to obtaining informed consent and within 28 days prior to study start may be used; such tests do not need to be repeated for screening. Patient must have stable liver tests prior to the first dose of study drug.

All screening evaluations must be completed and reviewed to confirm that patients meet all eligibility criteria before study start. The investigator will maintain a screening log to record details of all patients screened and to confirm eligibility or record reasons for screening failure, as applicable.

Patients in Cohort 1 will not contribute to Phase II; however, they will be followed-up until EOS. In Randomized Phase II, patients will be randomized in a 2:1 ratio to receive

T-DM1 or the combination of T-DM1 and capecitabine prior to receiving the first dose of study medication.

The IxRS will be available 24 hours a day, 7 days a week. Detailed instructions regarding the IxRS will be provided to each study center. The screening numbers are to be allocated according to the specification document agreed with the IxRS provider.

Please see Appendix 1 for the schedule of screening assessments.

# 4.5.2.2 Assessments during Treatment

#### For Patients with mBC

Scheduled study visits are based on a q3w cycle, with Cycle 1 beginning at Day 1. All visits must occur within ± 3 business days from the scheduled date, unless otherwise noted in the schedule of assessments. All assessments will be performed on the day of the specified visit unless a time window is specified. Assessments scheduled on the day of study treatment administration should be performed prior to study treatment administration unless otherwise noted. If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend, it should be performed on the nearest following date (i.e., within 3 business days).

Local laboratory assessments scheduled for Day 1 of all cycles must be performed within 72 hours prior to study treatment administration unless otherwise specified. Results of local laboratory assessments must be reviewed and the review documented prior to study treatment administration.

Please see Appendix 1 for the schedule of treatment period assessments.

#### For Patients with mGC

Scheduled study visits are based on a qw cycle, with Cycle 1 beginning at Day 1. All visits must occur within ± 3 business days from the scheduled date, unless otherwise noted in the schedule of assessments. All assessments will be performed on the day of the specified visit unless a time window is specified. Assessments scheduled on the day of study treatment administration should be performed prior to study treatment administration unless otherwise noted. If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend, it should be performed on the nearest following date (i.e., within 3 business days).

Local laboratory assessments scheduled for Day 1 of all cycles must be performed within 72 hours prior to study treatment administration unless otherwise specified. Results of local laboratory assessments must be reviewed and the review documented prior to study treatment administration.

Please see Appendix 1 for the schedule of treatment period assessments.

# 4.5.2.3 Assessments at Study Completion/Early Termination Visit

Patients may remain on study treatment until disease progression as assessed by the investigator, intolerable toxicity, or until the patient wishes to withdraw from study treatment. Patients who discontinue study treatment will be followed-up until EOS and will be asked to return to the clinic approximately 28–42 days after the last study treatment administration for the safety follow-up visit.

Please see Appendix 1 for assessments to be performed at the safety followup visit.

# 4.5.2.4 Follow-up Assessments

After the Study Treatment Discontinuation Visit, all patients (regardless of reason for discontinuation) will have anti-cancer therapies recorded and will be followed for all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up, or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.

Patients who discontinue study drugs for any reason other than disease progression or withdrawal of consent (e.g., an AE) will continue to be followed until the development of disease progression, consent withdrawal, lost to follow-up, or beginning of another anti-cancer therapy.

After the study completion/early termination visit, AEs should be followed as outlined in Section 5.5 and 5.6.

Please see Appendix 1 for the schedule of follow-up assessments.

#### 4.5.2.5 Assessments at Unplanned Visits

In case unplanned visits are required, electronic Case Report Form (eCRF) pages will be available to report the information collected during those visits.

# 4.6 PATIENT, STUDY, AND SITE DISCONTINUATION

#### 4.6.1 PATIENT DISCONTINUATION

Patients have the right to withdraw from the study at any time for any reason. The investigator has the right to discontinue a patient from study treatment or from the study for any medical condition that the investigator determines may jeopardize the patient's safety if he or she continues in the study, for reasons of non-compliance (e.g., missed doses, visits), if the patient becomes pregnant, or if the investigator determines it is in the best interest of the patient.

Patients must be withdrawn from study treatment if they become pregnant or experience disease progression defined using RECIST v. 1.1 Appendix 3. The exception to this is patients who develop isolated progression in the brain as described in Appendix 3.

Details of discontinuation due to toxicity are given in Section 5.1.

Other reasons for patient discontinuation may include, but are not limited to, the following:

- Pregnancy
- Non-compliance
- Investigator decision based on the patient's best interest

#### Patient decision

Patients who discontinue from study treatment prematurely for any of the above reasons will continue to be followed according to Section 4.5.2.4 "Follow-Up Assessments". The primary reason for discontinuation must be recorded on the appropriate eCRF page.

#### 4.6.2 STUDY DISCONTINUATION

Section 3.1.1 describes the EOS definition and discontinuation of study. Prior to that, the Sponsor has the right to terminate this study at any time. Reasons for terminating the study may include, but are not limited to, the following:

- The incidence or severity of AEs in this or other studies indicates a potential health hazard to patients
- Patient enrollment is unsatisfactory
- Data recording is inaccurate or incomplete

# 5. ASSESSMENT OF SAFETY

Overall safety will be assessed on an ongoing basis during the conduct of the study.

### 5.1 SAFETY PLAN

The safety plan for patients receiving trastuzumab emtansine is based on the toxicities of trastuzumab emtansine observed in nonclinical studies; the toxicities related to its components (trastuzumab and maytansine, the parent drug of DM1) observed in clinical studies; and the clinical experience with this molecule in completed and ongoing studies. Please refer to the trastuzumab emtansine and capecitabine (Xeloda®) Investigator`s Brochures for the most recent information.

All patients will be monitored closely for toxicity. The important safety issues anticipated in this trial, as well as measures intended to avoid or minimize such toxicities, are outlined in the following sections.

# 5.1.1 RISKS ASSOCIATED WITH TRASTUZUMAB EMTANSINE

Full details regarding the clinical safety of trastuzumab emtansine are presented in Sections 5 and 6 of the Investigator's Brochure.

# 5.1.1.1 Cardiotoxicity

Patients treated with trastuzumab emtansine are at increased risk of developing left ventricular dysfunction. LVEF < 40% has been observed in patients treated with trastuzumab emtansine. Patients without significant cardiac history and with an LVEF ≥ 50% determined by ECHO or MUGA scan are eligible for study participation. LVEF will be monitored at screening and regularly throughout the study until the assessment at the safety follow-up visit. Patients with symptomatic cardiac dysfunction will be discontinued from study treatment. Asymptomatic LVEF declines will be handled as per the

algorithm shown in Figure 6. Treatment with trastuzumab emtansine has not been studied in patients with LVEF < 50%.

# 5.1.1.2 Hematologic Toxicity (Thrombocytopenia)

Thrombocytopenia, or decreased platelet counts, was reported in patients in clinical trials of trastuzumab emtansine. The majority of these patients had Grade 1 or 2 events ( $\geq 50,000/\text{mm}^3$ ), with the nadir occurring by Day 8 and generally improving to Grade 0 or 1 ( $\geq 75,000/\text{mm}^3$ ) by the next scheduled dose. In clinical trials, the incidence and severity of thrombocytopenia were higher in Asian patients. Severe cases of both non-fatal and fatal hemorrhagic events including central nervous system hemorrhage have been reported in clinical trials with trastuzumab emtansine; these events were independent of the patients' ethnicity. In some of the observed cases the patients were also receiving anti-coagulation therapy. The need for platelet transfusions has been reported.

Patients with thrombocytopenia and on anti-coagulant treatment have to be monitored closely during treatment with trastuzumab emtansine. Platelet counts will be monitored prior to each trastuzumab emtansine dose.

Use of erythropoiesis-stimulating agents will be allowed as consistent with prescribing guidelines. Transfusion of red blood cells and/or platelets will be allowed according to and at the discretion of the treating physician.

# 5.1.1.3 Hepatotoxicity

Hepatotoxicity, predominantly in the form of asymptomatic increases in the concentrations of serum transaminases (Grade 1 – 4 transaminitis), has been observed in patients while on treatment with trastuzumab emtansine in clinical trials. Transaminase elevations were generally transient. The incidence of increased AST was substantially higher than that for ALT. The proportion of patients with Grade 1 or 2 increases in transaminases increased with successive cycles, suggesting a modest cumulative effect of trastuzumab emtansine on transaminases; however, no increase over time in the proportion of Grade 3 abnormalities was observed. Patients with elevated transaminases improved to Grade 1 or normal within 30 days of the last dose of trastuzumab emtansine in the majority of the patients.

Rare cases of severe hepatotoxicity, including death due to drug-induced liver injury and associated hepatic encephalopathy, have been observed in patients treated with trastuzumab emtansine. While there is evidence of drug-induced liver toxicity (predominantly in the form of asymptomatic increases in the concentrations of serum transaminases) in patients treated with trastuzumab emtansine, its potential to cause acute severe liver injury with clinically meaningful changes in liver function is unclear as the observed cases of acute liver injury were confounded by concomitant medications with known hepatotoxic potential and/or underlying conditions. Nevertheless, a contributory role of trastuzumab emtansine in these cases cannot be excluded. Therefore, acute severe liver injury (Hy's law) remains an important potential

risk with trastuzumab emtansine. A Hy's law case has the following components:

- Aminotransferase enzymes (ALT/AST) greater than 3 × ULN with concurrent elevation of serum total bilirubin to > 2 × ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)
- No other reason can be found to explain the combination of increased aminotransferases and serum total bilirubin, such as viral hepatitis A, B, or C, pre-existing or acute liver disease, or another drug capable of causing the observed injury
- The finding should be serious as shown by gross jaundice, clinical disability, need for hospital care, and be at least probably drug-induced (by trastuzumab emtansine)

Trastuzumab emtansine treatment in patients with serum transaminases  $> 3 \times \text{ULN}$  and concomitant total bilirubin  $> 2 \times \text{ULN}$  should be permanently discontinued.

Patients must have adequate and stable liver function: hepatic transaminases (AST/ALT) and total bilirubin must be within acceptable range, as defined in the protocol, within 4 weeks prior to the first dose of trastuzumab emtansine. Liver function will be monitored prior to each trastuzumab emtansine dose.

Cases of nodular regenerative hyperplasia (NRH) of the liver have been identified from liver biopsies in patients treated with trastuzumab emtansine and presenting with signs and symptoms of portal hypertension. NRH was also observed in one fatal case of hepatic failure. NRH is a rare liver condition characterized by widespread benign transformation of hepatic parenchyma into small regenerative nodules; NRH may lead to non-cirrhotic portal hypertension. Diagnosis of NRH can only be confirmed by histopathology.

NRH should be considered in patients who develop clinical symptoms of portal hypertension and/or a cirrhosis-like pattern seen on CT scan of the liver but with normal transaminases and no other manifestations of cirrhosis or liver failure following long-term treatment with trastuzumab emtansine. Upon diagnosis of NRH, trastuzumab emtansine treatment must be permanently discontinued.

# 5.1.1.4 Pulmonary Toxicity

Cases of interstitial lung disease (ILD), including pneumonitis, some leading to acute respiratory distress syndrome or fatal outcome, have been reported in clinical trials with trastuzumab emtansine. Signs and symptoms include dyspnea, cough, fatigue, and pulmonary infiltrates. These events may or may not occur as sequelae of infusion reactions. Treatment has included administration of steroids and oxygen, and study drug discontinuation. Patients with dyspnea at rest due to complications of advanced malignancy and comorbidities may be at increased risk of pulmonary events.

Treatment with trastuzumab emtansine has to be permanently discontinued in patients who are diagnosed with ILD or pneumonitis.

# 5.1.1.5 Infusion-related Reactions/Hypersensitivity

Infusion-related reactions characterized by one or more of the following symptoms, flushing, chills, pyrexia, dyspnea, hypotension, wheezing, bronchospasm, and tachycardia may occur with the administration of monoclonal antibodies and have been reported with trastuzumab emtansine. In general, these symptoms were not severe. In most patients, these reactions resolved over the course of several hours to a day after the infusion was terminated. Patients should be observed closely for infusion-related reactions, especially during the first infusion.

Patients should be observed closely for hypersensitivity. Serious, allergic/anaphylactic-like reactions have been observed in clinical trials with treatment of trastuzumab emtansine. Administration of trastuzumab emtansine will be performed in a setting with access to emergency facilities and staff who are trained to monitor and respond to medical emergencies. Patients will be observed closely for infusion-related/hypersensitivity during and after each trastuzumab emtansine infusion for a minimum of 90 minutes after the first infusion and for a minimum of 30 minutes after subsequent infusions in the absence of infusion-related AEs. Pre-medication is allowed according to standard practice guidelines. In the event of a true hypersensitivity reaction (in which severity of reaction increases with subsequent infusions), trastuzumab emtansine treatment must be permanently discontinued. Patients who experience a Grade  $\geq$  3 allergic reaction or acute respiratory distress syndrome will be discontinued from study treatment.

# 5.1.1.6 Neurotoxicity

DM1, an anti-microtubule agent, can potentially cause peripheral neuropathy. Peripheral neuropathy, mainly Grade 1 and predominantly sensory, has been reported in clinical trials of trastuzumab emtansine. Treatment with trastuzumab emtansine should be temporarily discontinued in patients experiencing Grade 3 or 4 peripheral neuropathy until symptoms resolve or improve to  $\leq$  Grade 2. Patients should be examined for signs of peripheral neuropathy prior to each dose of trastuzumab emtansine. Patients who experience Grade  $\geq$  3 neurotoxicity in the form of peripheral neuropathy that does not resolve to Grade  $\leq$  2 within 42 days after last dose received will be discontinued from study treatment.

#### 5.1.1.7 Extravasation

In trastuzumab emtansine clinical studies, reactions secondary to extravasation have been observed. These reactions were usually mild and comprised erythema, tenderness, skin irritation, pain, or swelling at the infusion site. Rare reports of more severe events such as cellulitis, pain (tenderness and burning sensation), and skin irritation have been received as part of the continuing surveillance of trastuzumab emtansine safety. These reactions have been observed more frequently within 24 hours of infusion. Specific treatment for trastuzumab emtansine extravasation is unknown at this

Study MO28230

time. The infusion site should be closely monitored for possible subcutaneous infiltration during drug administration.

#### 5.1.1.8 Trastuzumab Emtansine Dose Modification

Trastuzumab emtansine dose modifications are described in Section 5.1.5.1.

#### 5.1.2 RISKS ASSOCIATED WITH CAPECITABINE

Patients treated with capecitabine should be carefully monitored for toxicity. Most AEs are reversible and do not require permanent discontinuation of therapy (please refer to the Xeloda<sup>®</sup> Investigator`s Brochure for more information).

The spectrum of cardiotoxicity observed with capecitabine is similar to that of other fluorinated pyrimidines. This includes myocardial infarction, angina, dysrhythmias, cardiac arrest, cardiac failure and electrocardiographic changes. These AEs may be more common in patients with a prior history of coronary artery disease.

A rare, unexpected, severe toxicity (e.g. stomatitis, diarrhea, neutropenia, and neurotoxicity) associated with 5-FU has been attributed to deficiency of DPD activity. Therefore, a link between decreased levels of DPD and increased, potentially fatal, toxic effects of 5-FU cannot be excluded.

Capecitabine can induce hand-foot syndrome (palmar-plantar erythrodysesthesia or chemotherapy-induced acral erythema), which is a cutaneous toxicity. For patients receiving capecitabine monotherapy in the metastatic setting, the median time to onset was 79 days (range 11–360 days), with a severity range of Grades 1 to 3. Grade 1 hand-foot syndrome is defined by numbness, dysesthesia/paresthesia, tingling or erythema of the hands and/or feet and/or discomfort which does not disrupt normal activities. Grade 2 is defined as painful erythema and swelling of the hands and/or feet and/or discomfort affecting the patient's activities of daily living (ADL). Grade 3 is defined as moist desquamation, ulceration, blistering or severe pain of the hands and/or feet and/or severe discomfort that causes the patient to be unable to work or perform ADL. If Grade 2 or 3 hand-foot syndrome occurs, administration of capecitabine should be interrupted until the event resolves or decreases in intensity to Grade 1. Following Grade 3 hand-foot syndrome, subsequent doses of capecitabine should be decreased.

Capecitabine can induce hyperbilirubinemia. Administration of capecitabine should be interrupted if treatment-related elevations in bilirubin of  $> 3.0 \times ULN$  or treatment-related elevations in hepatic aminotransferases (ALT/AST) of Grade  $\geq 2$  occur.

# 5.1.3 RISKS ASSOCIATED WITH TRASTUZUMAB EMTANSINE AND CAPECITABINE COMBINATION

DLTs for the combination of trastuzumab emtansine and capecitabine will be observed during Cycle 1 (Day 1–21) of this study. The combination treatment must be considered as a new treatment during Cycle 1, and no individual

dose reduction will be allowed; the general DLT rules will be used instead. Interruptions can be made due to toxicities considered by the investigator to be related to capecitabine. Grade 2–4 toxicities should be interrupted until resolved to Grade 0–1. For Grade 4 toxicities, consideration to discontinue treatment with capecitabine will be made with the adjudication of the SC.

#### 5.1.4 DEFINITION OF DOSE-LIMITING TOXICITY

DLT toxicities will be observed during Cycle 1 (Day 1–21). Please refer to Xeloda<sup>®</sup> SmPC for recommendations on dose reduction.

# **Definition of DLT:**

# **Hematologic**

- Uncomplicated thrombocytopenia Grade 4 which does not recover to ≥ 75,000/MI before Day 21
- 2. Thrombocytopenia (any grade) complicated with clinically significant bleeding requiring medical intervention such as: platelet transfusion, cauterization, patients with epistaxis Grade 1 or 2 may have cauterization and this should not be consider as DLT etc.
- 3. Neutropenia Grade 4 lasting > 7 consecutive days
- 4. Febrile neutropenia with an ANC of < 1,000 cells/mm<sup>3</sup>

#### Non-hematologic

- 5. Diarrhea Grade ≥ 3 which does not decrease to ≤ Grade 2 after 24 hours of starting recommended anti-diarrheal treatment
- 6. Hand-foot syndrome Grade ≥ 3
- 7. Any other treatment-related toxicity ≥ Grade 3 prohibiting the start of the 2nd cycle on Day 22 (3 weeks cycle length plus 1 day)

NOTE: If a Grade 2 event requires a dose delay, it will not be considered as DLT. However, if the toxicity does not resolve to Grade 1 or baseline by Day 42, this requires discontinuation and will be considered as DLT.

- 8. Grade 2 toxicity requiring interruption of treatment for > 14 days NOTE: Patients experiencing ≥ Grade 3 hand-foot syndrome or diarrhea or mucositis or febrile neutropenia with ANC < 500 cells/mm³ during Cycle 1 must be tested for DPD deficiency (central laboratory will be appointed). The SC will adjudicate in cases of DLTs that are not covered by the existing DLT criteria.
- 9. Having taken < 14 full doses of capecitabine due to toxicity
- Patient not able to receive 100% of the dose level going into Cycle 2, Day 1

# 5.1.5 MANAGEMENT OF SPECIFIC ADVERSE EVENTS

#### 5.1.5.1 Trastuzumab Emtansine Dose Modification

Patients should be assessed for toxicity prior to each dose; dosing will occur only if the clinical assessment and laboratory test values are acceptable.

Dose delays and reductions are designed to maximize treatment for those who derive clinical benefit from treatment while ensuring patient safety. Dose delays for trastuzumab emtansine-related toxicity other than those specified below (i.e., infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, cardiotoxicity, and ILD or pneumonitis) are as follows:

- If significant trastuzumab emtansine-related toxicities (other than infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, and cardiotoxicity) have not recovered to Grade 1 or baseline, the next scheduled dose may be delayed for up to 42 days from the last dose received. "Significant" and "related" will be based on the judgment of the investigator (in consultation with the Sponsor's Medical Monitor or designee when appropriate). For example, alopecia even if considered related would most likely not be considered to be significant. Fatigue may or may not be considered either related or significant.
- In general, when the significant and related toxicity (or any other toxicity that the investigator chooses to delay dosing for) resolves to Grade 1 or baseline, the patient may resume trastuzumab emtansine if the delay has not exceeded 42 days from the last received dose. Patients should be reevaluated qw during the delay, whenever possible. If dosing resumes, the patient may receive trastuzumab emtansine either at the same dose level as before or at one dose level lower (see Table 2 and Table 3), at the discretion of the investigator. Subsequent cycles should remain the same (q3w or qw), and patients should be assessed for toxicity.
- If a patient requires a dose reduction, dosing will be reduced by one dose level, per Table 2 or Table 3. No dose re-escalation will be allowed.
- If toxicity does not resolve within 42 days from the last dose received, the patient will be discontinued from study treatment and will be followed for disease progression and survival outcome as described in Section 5.5.
- Patients who experience a Grade 3 or 4 hematologic event should be checked at least weekly for recovery. If values do not recover to baseline or Grade ≤ 1 within 42 days from the last dose received, the patient will be discontinued from study treatment.

Table 2 Dose Reduction for Trastuzumab Emtansine (Patients with mBC)

| Dose Level | q3w Schedule |
|---------------------------------------|---------------------|
| 0 | 3.6 mg/kg |
| - 1 | 3.0 mg/kg |
| - 2 | 2.4 mg/kg |
| Indication for further dose reduction | Off study treatment |

q3w = every 3 weeks

Table 3 Dose Reductions for Trastuzumab Emtansine (Patients with mGC)

| Dose Level | qw Schedule |
|---------------------------------------|-------------|
| 0 | 2.4 mg/kg |
| - 1 | 2.0 mg/kg |
| - 2 | Off study |
| Indication for further dose reduction | Off study |

qw = weekly

In case of toxicities requiring the discontinuation of T-DM1, the patient will be followed-up until the EOS.

Protocol requirements for specific toxicities are outlined below.

# 5.1.5.1.1 Trastuzumab Emtansine Dose Modification for Thrombocytopenia

Platelet counts should be obtained no less frequently than weekly to evaluate recovery whenever any of the events listed below occurs. If platelet counts do not recover to Grade ≤ 1 within 42 days from the last dose received, the patient will be discontinued from study treatment.

No re-escalation of the trastuzumab emtansine dose is allowed.

Note: although complete blood counts with platelets are required within 72 hours prior to study treatment administration at each cycle, the investigator may monitor platelet counts (or any other laboratory test) more frequently as clinically indicated.

In the event of decreased platelet count to Grade 3 ( $< 50,000/\text{mm}^3$ ), do not administer trastuzumab emtansine until platelet counts recover to Grade 1 ( $\ge 75,000/\text{mm}^3$ ), then treat at the same dose level.

Patients receiving trastuzumab emtansine who experience a first Grade 4 thrombocytopenia event may, after adequate recovery to a platelet count of


Grade  $\leq$  1 or baseline, continue treatment with trastuzumab emtansine at a dose of 3 mg/kg in subsequent treatment cycles. Patients at the 3 mg/kg dose level who experience a Grade 4 thrombocytopenia event may, after adequate recovery as defined above, continue treatment with trastuzumab emtansine at a dose of 2.4 mg/kg in subsequent treatment cycles. Patients who experience a Grade 4 thrombocytopenia event at the 2.4 mg/kg dose level will be discontinued from study treatment. A dose delay of up to 42 days from the patient's last dose received is permitted.

# 5.1.5.1.2 Trastuzumab Emtansine Dose Modification for Hepatotoxicity

# 5.1.5.1.2.1 Concurrent elevations of ALT/AST and bilirubin meeting Hy's Law laboratory criteria

Regardless of dose level, trastuzumab emtansine must be <u>permanently</u> <u>discontinued</u> in patients with ALT and/or AST > 3 × ULN and concurrent increase of total bilirubin to > 2 × ULN. All relevant hepatic laboratory tests performed (including AST, ALT, total bilirubin, alkaline phosphatase, activated partial thromboplastin time [aPTT], INR, and albumin) will be entered into the clinical database.

# 5.1.5.1.2.2 Nodular regenerative hyperplasia (NRH)

Trastuzumab emtansine must be permanently discontinued in patients who are diagnosed with NRH.

# 5.1.5.1.2.3 Transaminase elevations or bilirubin elevation requiring dose adjustment

Patients who experience a Grade 3 elevation of liver function should be checked twice weekly for the recovery of transaminases and/or total bilirubin. If a patient's transaminases and/or total bilirubin do not recover as per Table 4 and Table 5, within 42 days from the patient's last dose received, the patient will be discontinued from study treatment.

No re-escalation of the trastuzumab emtansine dose is allowed.

Table 4 and Table 5 describe the dose modification guidelines for increases in serum bilirubin and transaminases, respectively.

Table 4 Trastuzumab Emtansine Dose Modification: Total Serum Bilirubin

| Grade 2 | Grade 3 | Grade 4 |
|---|---|---|
| (> 1.5 to ≤ 3 × the ULN) | (> 3 to ≤ 10 × the ULN) | (> 10 × the ULN) |
| Do not administer T-DM1 until total bilirubin recovers to Grade ≤ 1, and then treat at the same dose level | Do not administer T-DM1 until total bilirubin recovers to Grade ≤ 1 and then reduce one dose level | Discontinue T-DM1 |

T-DM1 = trastuzumab emtansine; ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

Table 5 Trastuzumab Emtansine Dose Modification: Serum ALT or AST

| Grade 2 | Grade 3 | Grade 4 |
|------------------------|---------------------------|-------------------|
| (> 3 to ≤ 5 × the ULN) | (> 5 to ≤ 20 × the ULN) | (> 20 × the ULN) |
| Treat at the same dose | Do not administer T-DM1 | Discontinue T-DM1 |
| level | until AST/ALT recovers to | |
| | Grade ≤ 2, and then | |
| | reduce one dose level | |

ALT = alanine transaminase; AST = aspartate transaminase; T-DM1 = trastuzumab emtansine; ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

### 5.1.5.1.3 Trastuzumab Emtansine Dose Modification for Neurotoxicity

Patients receiving trastuzumab emtansine who experience Grade 3 or 4 peripheral neuropathy that does not resolve to Grade ≤ 2 within 42 days after the last dose received will be discontinued from study treatment.

# 5.1.5.1.4 Trastuzumab Emtansine Dose Modification for Cardiotoxicity

Patients without significant cardiac history and with a baseline LVEF ≥ 50% as determined by ECHO or MUGA scan are eligible for study participation. Ejection fractions will be monitored during the last week of Cycle 1, Cycle 3 and every third cycle thereafter until the assessment at the safety follow-up visit.

Figure 6 summarizes the management of trastuzumab emtansine on the basis of measured LVEF and changes in LVEF from baseline in patients. If the LVEF is reported as a range, the median of the range should be taken. If an investigator is concerned that an AE may be related to cardiac dysfunction, an
additional LVEF measurement may be performed. Trastuzumab emtansine will be discontinued in any patient who develops symptomatic CHF. CHF should be treated and monitored according to standard medical practice.

The decision to stop or continue trastuzumab emtansine should be based on the algorithm shown in Figure 6. Trastuzumab emtansine must be discontinued in all patients for whom a confirmed drop of LVEF to below 40% is documented (with a repeat assessment within 21 days). For patients whose LVEF drops to values between 40% and 45% with an absolute decrease in LVEF of ≥ 10% points from baseline, trastuzumab emtansine should be held. For these patients, the LVEF should be repeated in 21 days, and trastuzumab emtansine should be discontinued if the LVEF has not recovered to within 10% absolute difference below baseline. If clinically significant cardiac dysfunction or cardiac failure develops or persists or if significant medical management is required to maintain ejection fraction, the patient should be discontinued from study treatment.

Figure 6 Algorithm for Continuation and Discontinuation of
Trastuzumab Emtansine Based on Left Ventricular Ejection
Fraction Assessments in Patients



CHF = congestive heart failure; LVEF = left ventricular ejection fraction.

Note: LVEF assessment results must be reviewed before the next scheduled trastuzumab emtansine infusion.

- LVEF can be repeated within 21 days, and trastuzumab emtansine should be discontinued if LVEF < 40% is confirmed. Trastuzumab emtansine should be held while the repeat LVEF is obtained.
- After a second consecutive confirmatory result, trastuzumab emtansine should be discontinued if the LVEF is confirmed to be ≥ 10% points below baseline or if medical management was required to correct the LVEF.

# 5.1.5.1.5 Trastuzumab Emtansine Dose Modification/Management for Infusion-related Reactions, Hypersensitivity Reactions

Trastuzumab emtansine treatment should be interrupted in patients with severe infusion-related reactions. Trastuzumab emtansine treatment should be permanently discontinued in the event of life-threatening infusion-related reactions.

Infusion of trastuzumab emtansine should be interrupted for patients who develop dyspnea or clinically significant hypotension.

The infusion should be slowed to  $\leq 50\%$  or interrupted for patients who experience any other infusion-related symptoms. When the patient's symptoms have completely resolved, the infusion may be continued at  $\leq 50\%$  of the rate prior to the reaction and increased in 50% increments every 30 minutes as tolerated. Infusions may be restarted at the full rate during the next cycle.

Study MO28230

Patients who experience trastuzumab emtansine infusion-related temperature elevations to > 38.5°C and/or other infusion-related symptoms may be treated symptomatically with acetaminophen and/or diphenhydramine hydrochloride. Serious infusion-related events manifested by dyspnea, hypotension, wheezing, bronchospasm, tachycardia, reduced oxygen saturation, or respiratory distress should be managed with supportive care, such as oxygen, beta agonists, antihistamines, antipyretics, or corticosteroids at the investigator's discretion. Pre-medication with corticosteroids, antihistamines, and antipyretics may be used before subsequent infusions of trastuzumab emtansine at the investigator's discretion. Patients should be monitored until complete resolution of symptoms. In the event of a true hypersensitivity reaction (i.e., if the severity of reaction increases with subsequent infusions), trastuzumab emtansine treatment must be permanently discontinued. Patients who experience a Grade ≥ 3 hypersensitivity reaction or acute respiratory distress syndrome (ARDS) will be discontinued from the study.

Patients who experience a severe delayed infusion reaction will be discontinued from study treatment.

# 5.1.5.1.6 Trastuzumab Emtansine Dose Modification for Pulmonary Toxicity

Cases of ILD, including pneumonitis (including severe, life-threatening cases) and some leading to ARDS or fatal outcome have been reported with trastuzumab emtansine. Treatment with trastuzumab emtansine has to be permanently discontinued in patients who are diagnosed with ILD or pneumonitis.

# 5.1.5.1.7 Trastuzumab Emtansine Dose Modification for Extravasation

During the clinical development of T-DM1, reactions secondary to extravasation have been observed. These reactions were usually mild and comprised of erythema, tenderness, skin irritation, pain or swelling at the infusion site. Although T-DM1 is not considered as a vesicant, close monitoring of the infusion site for possible subcutaneous infiltration during drug administration is recommended.

# 5.1.5.2 Capecitabine Dosage Modification

# Phase I: Patients with mBC

The dose of capecitabine can be modified if considered appropriate by the investigator (please refer to the Xeloda<sup>®</sup> SmPC for recommendations).

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued in patients with mBC.

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

During the Randomized Phase II part of the study, the dose of capecitabine will be modified as per the Xeloda<sup>®</sup> SmPC.


In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued in patients with mBC.

# Phase I: Patients with mGC

The dose of capecitabine can be modified if considered appropriate by the investigator (please refer to Xeloda<sup>®</sup> SmPC for recommendations).

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued in patients with mGC.

# 5.2 SAFETY PARAMETERS AND DEFINITIONS

Safety assessments will consist of monitoring and recording protocol-defined AEs and SAEs; measurement of protocol-specified hematology, clinical chemistry, and urinalysis variables; measurement of protocol-specified vital signs; and other protocol-specified tests that are deemed critical to the safety evaluation of the study drug(s).

The Sponsor or its designee is responsible for reporting relevant SAEs to the Competent Authority, other applicable regulatory authorities, and participating investigators, in accordance with International Conference on Harmonisation (ICH) guidelines, Food and Drug Administration (FDA) regulations, European Clinical Trials Directive (Directive 2001/20/EC), and/or local regulatory requirements.

The Sponsor or its designee is responsible for reporting unexpected fatal or life-threatening events associated with the use of the study drug to the regulatory agencies and competent authorities by telephone or fax within 7 calendar days after being notified of the event. The Sponsor or its designee will report other relevant SAEs associated with the use of the study medication to the appropriate competent authorities (according to local guidelines), investigators, and central Institutional Review Boards/Ethics Committees (IRBs/ECs) by a written safety report within 15 calendar days of notification.

# 5.2.1 ADVERSE EVENTS

According to the ICH Guideline for Good Clinical Practice, an AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any of the following:

- Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
- Any new disease or exacerbation of an existing disease (a worsening in the character, frequency, or severity of a known condition), except as described in Section 5.3.5.7
- Recurrence of an intermittent medical condition (e.g., headache) not present at baseline

- Any deterioration in a laboratory value or other clinical test (e.g., ECG, X-ray) that is associated with symptoms or leads to a change in study treatment or concomitant treatment or discontinuation from study drug
- AEs that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment (e.g., screening invasive procedures such as biopsies)

# 5.2.2 SERIOUS ADVERSE EVENTS (IMMEDIATELY REPORTABLE TO THE SPONSOR)

A SAE is any AE that meets any of the following criteria:

- Fatal (i.e., the AE actually causes or leads to death)
- Life-threatening (i.e., the AE, in the view of the investigator, places the patient at immediate risk of death)

This does not include any AE that had it occurred in a more severe form or was allowed to continue might have caused death.

- Requires or prolongs inpatient hospitalization (see Section 5.3.5.8)
- Results in persistent or significant disability/incapacity (i.e., the AE results in substantial disruption of the patient's ability to conduct normal life functions)
- Congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug
- Significant medical event in the investigator's judgment (e.g., may jeopardize the patient or may require medical/surgical intervention to prevent one of the outcomes listed above)

The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an AE (rated as mild, moderate, or severe, or according to NCI CTCAE criteria; see Section 5.3.3); the event itself may be of relatively minor medical significance (such as severe headache without any further findings).

Severity and seriousness need to be independently assessed for each AE recorded on the eCRF.

SAEs are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2 for reporting instructions).

# 5.2.3 PROTOCOL-DEFINED EVENTS OF SPECIAL INTEREST/NON-SERIOUS EXPEDITED ADVERSE EVENTS

Non-serious AESIs are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2 for reporting instructions). AESIs for this study include the following:

Potential drug-induced liver injury

Study MO28230

Any potential case of drug-induced liver injury as assessed by laboratory criteria for Hy's law will be considered as a protocol-defined event of special interest and will need to be reported to the Sponsor expeditiously.

The following laboratory abnormalities define potential Hy's law cases:

AST and/or ALT elevations that are > 3 × ULN with concurrent elevation
of total bilirubin > 2 × ULN, except in patients with documented Gilbert's
syndrome. For patients with Gilbert's syndrome, elevation of direct
bilirubin > 2 × ULN should be used instead

Suspected transmission of an infectious agent by the study drug:

 Defined as any organism, virus, or infectious particle (e.g., prion protein transmitting transmissible spongiform encephalopathy), both pathogenic and non-pathogenic. A transmission of an infectious agent may be suspected from clinical symptoms or laboratory findings indicating an infection in a patient exposed to a medicinal product. This term ONLY applies when a contamination of the study drug is suspected, NOT for infections supported by the mode of action, e.g., immunosuppression.

#### 5.2.4 Pregnancy and Contraception

ICH M3 guidance requires precautions to be taken to minimize risk to fetus or embryo when including women of childbearing potential in clinical studies. These precautions include the use of highly effective contraceptive measures, excluding pregnancy at baseline (serum test), continued pregnancy monitoring, and continued pregnancy testing for up to 6 months following last dose of study drug (follow-up period based on PK considerations).

Trastuzumab, a component of trastuzumab emtansine, can cause fetal harm when administered to a pregnant woman; postmarketing case reports indicate that its use during pregnancy increases the risk for oligohydramnios during the second and third trimester. Trastuzumab has also been associated with fetal pulmonary hypoplasia, skeletal abnormalities, and neonatal death (see the Herceptin<sup>®</sup> Package Insert). There are no clinical studies of trastuzumab in pregnant women. Immunoglobulin G (IgG) is known to cross the placental barrier.

Therefore, trastuzumab emtansine should be not used during pregnancy. Women of childbearing potential (who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy) and men with partners of childbearing potential must agree to use a highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the patient and/or partner.

Methods of birth control which result in a low failure rate (i.e., < 1% per year) when used consistently and correctly are considered highly effective forms of contraception. The use of the following non-hormonal methods of contraception is acceptable:

 True abstinence, when this is the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, and symptothermal

- post ovulation methods) and withdrawal are not acceptable methods of contraception.
- Male sterilization (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female patients, the vasectomized male partner should be the sole partner.

Alternatively, use of two of the following effective forms of contraception is acceptable:

- Placement of intrauterine device (IUD) or intrauterine system (IUS).
   Consideration should be given to the type of device being used, as there are higher failure rates for certain types (e.g., steel or copper wire).
- Condom with spermicidal foam/gel/film/cream/suppository
- Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

The use of barrier contraceptives should always be supplemented with the use of a spermicide. The following should be noted:

- Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection.
- However, spermicides alone are ineffective at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

It should be noted that two forms of effective contraception are required. A double barrier method, defined as condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, is acceptable.

Contraception is not a requirement in the case of any of the following:

- The female patient or female partner of a male patient is considered not to be of childbearing potential: if she is postmenopausal, defined by amenorrhea of ≥ 12 months duration in a woman > 45 years old; or is ≥ 40 years of age and has had amenorrhea of ≥ 24 months duration; or has undergone surgical sterilization (hysterectomy and/or bilateral oophorectomy)
- The male patient or male partner of a female patient is surgically sterilized

For male patients with a female partner of childbearing potential, cooperation of female partner is required (i.e., use of two forms of contraception as stated above) during the study and for at least 6 months following the last dose of study treatment when a highly effective form of contraception is not appropriate.

Based on PK considerations, contraception must continue for the duration of study treatment and for at least 6 months after the last dose of study treatment.

A female patient who becomes pregnant during the study must be instructed to stop taking the study medication and immediately inform the investigator. The investigator should report all pregnancies within 24 hours to the Sponsor including the partners of male patients. The investigator should counsel the patient/partner, and discuss the risks of continuing with the pregnancy and the possible effects on the fetus. Monitoring of the patient/partner should continue until conclusion of the pregnancy. Pregnancies occurring up to 6 months after the completion of study medication must also be reported to the investigator. Please refer to Section 5.4.3 for reporting procedures.

It is not known whether trastuzumab or trastuzumab emtansine are excreted in human milk. Maternal IgG is excreted in milk and any of these monoclonal antibodies could harm infant growth and development; therefore, women should be advised to discontinue nursing during trastuzumab emtansine therapy and not to breastfeed for at least 6 months following the last dose of either study drug.

Experimental studies have reported that IgGs are present in both the preejaculate and the seminal plasma (Moldoveanu et al. 2005). To date, there
have been no clinical studies to assess the IgG profile in the pre-ejaculate and
seminal plasma in male patients receiving trastuzumab or trastuzumab
emtansine. Therefore, as a precaution male patients with female partners of
childbearing potential are required to use highly effective form of
contraception or use two forms of contraception as outlined above. Similarly,
vaginal absorption of trastuzumab emtansine is unknown and therefore male
patients with pregnant partners are required to use condoms for the duration
of the pregnancy, and then revert to contraceptive methods as outlined above.
This is to ensure that the fetus is not exposed to the study medication through
vaginal absorption. In addition, sperm or blood donation should not occur for
at least 6 months after the last dose of study treatment.

# 5.3 METHODS AND TIMING FOR CAPTURING AND ASSESSING SAFETY PARAMETERS

The investigator is responsible for ensuring that all AEs (see Section 5.2.1 for definition) are recorded on the AE eCRF and reported to the Sponsor in accordance with instructions provided in this section and in Sections 5.4, 5.5, and 5.6.

For each AE recorded on the AE eCRF, the investigator will make an assessment of seriousness (see Section 5.2.2, for seriousness criteria), severity (see Section 5.3.3), and causality (see Section 5.3.4).

# 5.3.1 ADVERSE EVENT REPORTING PERIOD

Investigators will seek information on AEs at each patient contact. All AEs, whether reported by the patient or noted by study personnel, will be recorded in the patient's medical record and on the AE eCRF.

After informed consent has been obtained but prior to initiation of study drug, only SAEs caused by a protocol-mandated intervention should be reported

(e.g., SAEs related to invasive procedures such as biopsies, medication washout, or no treatment run-in).

After initiation of study treatment, all AEs, regardless of relationship to study drug, will be reported until 30 days after the last administration of study drug or study discontinuation/termination, whichever is later. After this period, all SAEs and non-serious AESIs (regardless of causality) occurring to a patient after the treatment of that patient has ended should be reported to the Sponsor if the investigator becomes aware of them. The investigator is not required to actively monitor patients after the study has ended (see Section 5.6).

# 5.3.2 ELICITING ADVERSE EVENT INFORMATION

A consistent methodology of non-directive questioning should be adopted for eliciting AE information at all patient evaluation time points. Examples of non-directive questions include the following:

"How have you felt since your last clinic visit?"

"Have you had any new or changed health problems since you were last here?"

# 5.3.3 ASSESSMENT OF SEVERITY OF ADVERSE EVENTS

The AE grading (severity) scale found in the NCI CTCAE (v. 4.0) will be used for assessing AE severity (see Table 6).

Table 6 Adverse Event Severity Grading Scale

| | Severity | Alternate Description <sup>a</sup> |
|---|---|---|
| Grade | | |
| 1 | Mild (apply event-specific NCI CTCAE grading criteria) | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate (apply event-specific NCI CTCAE grading criteria) | Minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental ADL <sup>b</sup> |
| 3 | Severe (apply event-specific NCI CTCAE grading criteria) | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL <sup>c</sup> |
| 4 | Very severe, life-threatening,<br>or disabling (apply event-specific<br>NCI CTCAE grading criteria) | Life-threatening consequences; urgent intervention indicated |
| 5 | Death related to AE | |

ADL = activities of daily living; AE = adverse event; CTCAE = Common Terminology Criteria for Adverse Events; NCI = National Cancer Institute.

The NCI CTCAE v4.0 can be found at:

http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm#ctc 40

Note: Regardless of severity, some events may also meet regulatory seriousness criteria. Refer to definition of a serious AE (see Section 5.2.2).

- <sup>a</sup> Use these alternative definitions for Grade 1, 2, 3, and 4 events when the observed or reported AE is not in the NCI CTCAE listing.
- Instrumental ADL refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
- Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

# 5.3.4 ASSESSMENT OF CAUSALITY OF ADVERSE EVENTS

Investigators should use their knowledge of the patient, the circumstances surrounding the event, and an evaluation of any potential alternative causes to determine whether or not an AE is considered to be related to study drugs, indicating "yes" or "no" accordingly. To ensure consistency of causality assessments, investigators should apply the general guidelines outlined in Table 7.

#### **Guidance for Causal Attribution of Adverse Event/Serious** Table 7 **Adverse Event**

Is the AE/SAE suspected to be caused by the investigational product based on facts, evidence, science-based rationales, and clinical judgment?

YES There is a plausible temporal relationship between the onset of the AE and administration of the investigational product, and the AE cannot be readily explained by the patient's clinical state, intercurrent illness, or concomitant therapies; and/or the AE follows a known pattern of response to the investigational product; and/or the AE abates or resolves upon discontinuation of the investigational product or dose reduction and, if applicable, reappears upon re-challenge.

Investigators should apply facts, evidence, or rationales based on scientific principles and clinical judgment to support a causal/contributory association with an investigational product.

AEs will be considered related, unless they fulfill the criteria as specified below. NO

Evidence exists that the AE has an etiology other than the investigational product (e.g., pre-existing medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the AE has no plausible temporal relationship to administration of the investigational product (e.g., cancer diagnosed 2 days after first dose of study drug).

Note: The investigator's assessment of causality for individual AE reports is part of the study documentation process. Regardless of the "Yes" or "No" causality assessment for individual AE reports, the Sponsor will promptly evaluate all reported SAEs against cumulative product experience to identify and expeditiously communicate possible new safety findings to investigators and applicable regulatory authorities. Attribution of SAEs will be reviewed on an ongoing basis, and may be changed as additional clinical data emerges (e.g., reversibility of AE, new clinical findings in patient with AE, effects of retreatment, AEs in other patients).

In addition to assessing causality with respect to study drugs, investigators should also assess whether other factors (e.g., disease under study, concurrent illness, concomitant medication, or study procedure) may have caused the event, using similar guidance.

The investigator's assessment of causality for individual AE reports is part of the study documentation process. Regardless of the "Yes" or "No" causality assessment for individual AE reports, the Sponsor will promptly evaluate all reported serious AEs against cumulative product experience to identify and expeditiously communicate possible new safety findings to investigators and applicable regulatory authorities.

For patients receiving combination therapy, causality will be assessed individually for each protocol-mandated therapy.

#### 5.3.5 PROCEDURES FOR RECORDING ADVERSE EVENTS

Investigators should use correct medical terminology/concepts when recording AEs on the AE eCRF. Avoid colloquialisms and abbreviations.

There is one eCRF page for recording AEs or SAEs.

Only one AE term should be recorded in the event field on the AE eCRF.

# 5.3.5.1 Diagnosis *versus* Signs and Symptoms

# Infusion-related Reactions

AEs that occur during or within 24 hours after study drug infusion should be captured as individual signs and symptoms rather than a diagnosis of allergic reaction or infusion-related reaction. However, a diagnosis has to be captured as an AE if signs and symptoms constitute a diagnosis of allergic reaction/hypersensitivity or infusion-related reaction and are classified as SAEs; all such symptoms have to be described in the narrative (e.g., in the Additional Case Details field of the eCRF).

# **Other Adverse Events**

For AEs other than infusion-related reactions, a diagnosis (if known) should be recorded on the AE eCRF rather than individual signs and symptoms (e.g., record only liver failure or hepatitis rather than jaundice, asterixis, and elevated transaminases). However, if a constellation of signs and/or symptoms cannot be medically characterized as a single diagnosis or syndrome at the time of reporting, each individual event should be recorded on the AE eCRF. If a diagnosis is subsequently established, all previously reported AEs based on signs and symptoms should be nullified and replaced by one AE report based on the single diagnosis, with a starting date that corresponds to the starting date of the first symptom of the eventual diagnosis.

# 5.3.5.2 Adverse Events Occurring Secondary to Other Events

In general, AEs occurring secondary to other events (e.g., cascade events or clinical sequelae) should be identified by their primary cause. For example, if severe diarrhea is known to have resulted in dehydration, it is sufficient to record only diarrhea as an AE or SAE on the eCRF.

However, medically significant AEs occurring secondary to an initiating event that are separated in time should be recorded as independent events on the eCRF. For example, if a severe gastrointestinal hemorrhage leads to renal failure, both events should be recorded separately on the eCRF.

# 5.3.5.3 Persistent or Recurrent Adverse Events

A persistent AE is one that extends continuously, without resolution, between patient evaluation time points. Such events should only be recorded once on the AE eCRF. The initial severity of the event should be recorded, and the severity should be updated to reflect the most extreme severity any time the event worsens. If the event becomes serious, the AE eCRF should be updated to reflect this.

A recurrent AE is one that resolves between patient evaluation time points and subsequently recurs. Each recurrence of an AE should be recorded separately on the AE eCRF.

# 5.3.5.4 Abnormal Laboratory Values

Only clinically significant laboratory abnormalities that require active management will be recorded as AEs or SAEs on the eCRF (e.g., abnormalities that require study drug dose modification, discontinuation of study treatment, more frequent follow-up assessments, further diagnostic investigation, etc.).

If the clinically significant laboratory abnormality is a sign of a disease or syndrome (e.g., alkaline phosphatase and bilirubin 5 × ULN of normal associated with cholecystitis), only the diagnosis (e.g., cholecystitis) needs to be recorded on the AE eCRF.

If the clinically significant laboratory abnormality is not a sign of a disease or syndrome, the abnormality itself should be recorded as an AE or SAE on the eCRF. If the laboratory abnormality can be characterized by a precise clinical term, the clinical term should be recorded as the AE or SAE. For example, an elevated serum potassium level of 7.0 mEq/L should be recorded as "hyperkalemia."

Observations of the same clinically significant laboratory abnormality from visit to visit should not be repeatedly recorded as AEs or SAEs on the eCRF, unless their severity, seriousness, or etiology changes.

# 5.3.5.5 Deaths

Deaths that occur during the protocol-specified AE reporting period (see Section 5.3.1), that are attributed by the investigator solely to progression of mBC or mGC should be recorded only on the Study Completion/Early Discontinuation eCRF. All other on-study deaths, regardless of relationship to study drug, must be recorded on the AE eCRF and immediately reported to the Sponsor (see Section 5.4.2). An independent monitoring committee will monitor the frequency of death from all causes.

Death should be considered an outcome and not a distinct event. The event or condition that caused or contributed to the fatal outcome should be recorded as the single medical concept on the AE eCRF. Generally, only one such event should be reported. If the cause of death is unknown and cannot be ascertained at the time of reporting, "unexplained death" should be recorded on the AE eCRF. If the cause of death later becomes available (e.g., after autopsy), "unexplained death" should be replaced by the established cause of death.

During post-study survival follow-up, deaths attributed to progression of mBC or mGC should be recorded only on the Survival eCRF.

# **5.3.5.6** Pre-Existing Medical Conditions

A pre-existing medical condition is one that is present at the start of this study. Such conditions should be recorded on the Medical and Surgical History eCRF.

A pre-existing medical condition should be recorded as an AE <u>only</u> if the frequency, severity, or character of the condition worsens during the study. When recording such events on the AE eCRF, it is important to convey the concept that the pre-existing condition has changed by including applicable descriptors (e.g., "more frequent headaches").

# 5.3.5.7 Lack of Efficacy or Clinical Worsening

Events that are clearly consistent with the expected pattern of progression of mBC or mGC should not be recorded as AEs. These data will be captured as efficacy assessment data only. In most cases, the expected pattern of progression will be based on the RECIST criteria. In rare cases, the determination of clinical progression will be based on symptomatic deterioration. However, every effort should be made to document progression using objective criteria. If there is any uncertainty as to whether an event is due to disease progression, it should be reported as an AE.

# 5.3.5.8 Hospitalization or Prolonged Hospitalization

Any AE that results in hospitalization or prolonged hospitalization should be documented and reported as a SAE unless specifically instructed otherwise in this protocol.

There are some hospitalization scenarios that do not require reporting as an SAE when there is no occurrence of an AE. These scenarios include a planned hospitalization or prolonged hospitalization to:

- Perform an efficacy measurement for the study
- Undergo a diagnostic or elective surgical procedure for a pre-existing medical condition that has not changed
- Receive scheduled therapy for the target disease of the study

# 5.4 IMMEDIATE REPORTING REQUIREMENTS FROM INVESTIGATOR TO THE SPONSOR

Certain events require immediate reporting to allow the Sponsor to take appropriate measures to address potential new risks in a clinical trial. The investigator must report such events to the Sponsor immediately; under no circumstances should reporting take place more than 24 hours after the investigator learns of the event. The following is a list of events that the investigator must report to the Sponsor within 24 hours after learning of the event, regardless of relationship to study drug:

- SAEs
- Non-serious AESIs
- Pregnancies

The investigator must report new significant follow-up information for these events to the Sponsor immediately (i.e., no more than 24 hours) after becoming aware of the information. New significant information includes the following:

Trastuzumab Emtansine 279 RO5304020 Study MO28230

- New signs or symptoms or a change in the diagnosis
- Significant new diagnostic test results
- Change in causality based on new information
- Change in the event's outcome, including recovery
- Additional narrative information on the clinical course of the event

Investigators must also comply with local requirements for reporting SAEs to the local health authority and Institutional Review Board/Ethics Committee (IRB/EC).

# 5.4.1 EMERGENCY MEDICAL CONTACTS

# MEDICAL MONITOR (SPONSOR'S MEDICAL RESPONSIBLE) CONTACT INFORMATION

To ensure the safety of study patients, an Emergency Medical Call Center Help Desk will access the Sponsor Medical Emergency List, escalate emergency medical calls, provide medical translation service (if necessary), connect the investigator with a Sponsor Medical Monitor, and track all calls. The Emergency Medical Call Center Help Desk will be available 24 hours per day, 7 days per week. Toll-free numbers for the Help Desk and Medical Monitor contact information will be distributed to all investigators (see "Protocol Administrative and Contact Information and List of Investigators").

# 5.4.2 REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS AND NON-SERIOUS ADVERSE EVENTS OF SPECIAL INTEREST

For reports of SAEs and non-serious AESIs, investigators should record all case details that can be gathered immediately (i.e., no more than 24 hours) on the AE eCRF and submit the report via the electronic data capture (EDC) system. A report will be generated and sent to the Sponsor Safety Risk Management by the EDC system.

In the event that the EDC system is unavailable, a paper SAE/Non-Serious AE of Special Interest CRF and Fax Coversheet should be completed and faxed to the Sponsor Safety Risk Management or its designee immediately (i.e., no more than 24 hours) after learning of the event, using the fax numbers provided to investigators (see "Protocol Administrative and Contact Information & List of Investigators"). Once the EDC system is available, all information will need to be entered and submitted via the EDC system.

# 5.4.3 REPORTING REQUIREMENTS FOR PREGNANCIES

# **5.4.3.1** Pregnancies in Female Patients

Female patients of childbearing potential will be instructed to immediately inform the investigator if they become pregnant during the study or within 6 months after the last dose of study drug. A Pregnancy Report eCRF should be completed by the investigator immediately (i.e., no more than 24 hours)

after learning of the pregnancy and submitted via the EDC system. A Pregnancy Report will automatically be generated and sent to the Sponsor Safety Risk Management. Pregnancy should not be recorded on the AE eCRF. The investigator should have the patient discontinue the study drug and discuss with the patient the risks of the pregnancy and the possible effects on the fetus. Monitoring of the patient should continue until conclusion of the pregnancy.

In the event that the EDC system is unavailable, a Pregnancy Report worksheet and Pregnancy Fax Coversheet should be completed and faxed to the Sponsor Safety Risk Management or its designee immediately (i.e., no more than 24 hours) after learning of the pregnancy, using the fax numbers provided to investigators (see "Protocol Administrative and Contact Information & List of Investigators").

# 5.4.3.2 Pregnancies in Female Partners of Male Patients

Male patients will be instructed through the Informed Consent Form to immediately inform the investigator if their partner becomes pregnant during the study or within 6 months after the last dose of study drug. A Pregnancy Report eCRF should be completed by the investigator immediately (i.e., no more than 24 hours) after learning of the pregnancy and submitted via the EDC system. Attempts should be made to collect and report details of the course and outcome of any pregnancy in the partner of a male patient exposed to study drug. The pregnant partner will need to sign an Authorization for Use and Disclosure of Pregnancy Health Information to allow for follow-up on her pregnancy. Once the authorization has been signed, the investigator will update the Pregnancy Report eCRF with additional information on the course and outcome of the pregnancy. An investigator who is contacted by the male patient or his pregnant partner may provide information on the risks of the pregnancy and the possible effects on the fetus, to support an informed decision in cooperation with the treating physician and/or obstetrician.

In the event that the EDC system is unavailable, follow reporting instructions provided in Section 5.4.3.1.

# 5.4.3.3 Abortions

Any spontaneous abortion should be classified as an SAE (as the Sponsor considers spontaneous abortions to be medically significant events), recorded on the AE eCRF, and reported to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2).

# 5.4.3.4 Congenital Anomalies/Birth Defects

Any congenital anomaly/birth defect in a child born to a female patient or female partner of a male patient exposed to study drug should be classified as an SAE, recorded on the AE eCRF, and reported to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2).

# 5.5 FOLLOW-UP OF PATIENTS AFTER ADVERSE EVENTS

# 5.5.1 INVESTIGATOR FOLLOW-UP

The investigator should follow all unresolved AEs and until the events are resolved or stabilized, the patient is lost to follow-up, or it has been determined that the study treatment or participation is not the cause of the AE/SAE. Resolution of AEs and SAEs (with dates) should be documented on the AE eCRF and in the patient's medical record to facilitate source data verification (SDV).

All pregnancies reported during the study should be followed until pregnancy outcome. If the EDC system is not available at the time of pregnancy outcome, follow reporting instructions provided in Section 5.4.3.1.

# 5.5.2 Sponsor Follow-up

For SAEs, non-serious AESIs, and pregnancies, the Sponsor or a designee may follow-up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details and outcome information (e.g., from hospital discharge summaries, consultant reports, autopsy reports) in order to perform an independent medical assessment of the reported case.

# 5.6 POST-STUDY ADVERSE EVENTS

At the study completion/early termination visit, the investigator should instruct each patient to report to the investigator any subsequent AEs that could be related or not related to the drug under observation.

The investigator should notify the Sponsor of any death, SAE or AESI occurring at any time after a patient has discontinued study participation. The Sponsor should also be notified if the investigator becomes aware of the development of cancer or a congenital anomaly/birth defect in a subsequently conceived offspring of a patient that participated in this study.

The investigator does not need to actively monitor patients for AEs once the trial has ended. The investigator should report the event directly to Roche Safety Risk Management via telephone or via facsimile using the Roche Clinical Trial (SAE) Reporting Form.

# 5.7 EXPEDITED REPORTING TO HEALTH AUTHORITIES, INVESTIGATORS, INSTITUTIONAL REVIEW BOARDS, AND ETHICS COMMITTEES

To determine reporting requirements for single AE cases, the Sponsor will assess the expectedness of these events using the following reference documents:

Trastuzumab emtansine and capecitabine Investigator's Brochures

The Sponsor will compare the severity of each event and the cumulative event frequency reported for the study with the severity and frequency reported in the applicable reference document.

Reporting requirements will also be based on the investigator's assessment of causality and seriousness, with allowance for upgrading by the Sponsor as needed.

The iDMC will closely monitor the incidence of these expected events during the study. An aggregate report of any clinically relevant imbalances that do not favor the test product will be submitted to health authorities.

#### 6. STATISTICAL CONSIDERATIONS AND ANALYSIS PLAN

# Phase I: Patients with mBC:

Enrollment into Cohort 1, patients with HER2-positive mBC, will open first.

Enrolled patients will receive study drug until Investigator-assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician, or study termination by the Sponsor.

Randomized Phase II: Exploration of Efficacy and Safety in mBC Patients randomized in Phase II will receive study drug until Investigator-assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician, or study termination by the Sponsor.

The final analysis of Randomized Phase II part of this study for ORR will be performed at the EOS (defined in Section 3.2).

# Phase I: Patients with mGC:

Once MTD is established for Cohort 1, enrollment of patients with HER2positive and locally advanced or mGC into Cohort 2 will be opened.

Enrolled patients will receive study drug until Investigator-assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician, or study termination by the Sponsor.

#### 6.1 **DETERMINATION OF SAMPLE SIZE**

# Sample Size for Phase I: mBC

This part will be based on a classical 3 plus 3 Phase I design. A minimum of 6 and up to 18 patients will be enrolled into Cohort 1. There is no formal sample size estimation for this part.

# Sample Size for Randomized Phase II: Exploration of Efficacy and Safety in mBC

Approximately 117 patients (78 patients in the combination of T-DM1 and capecitabine respective 39 patients in TDM1 treatment group), including a 10% withdrawal rate, will be randomized with a 2:1 ratio to the combination of T-DM1 and capecitabine or T-DM1.

Point estimates and 95% Clopper-Pearson exact CIs are tabulated for a range of possible BOR outcomes for both treatment groups in Table 8.

Table 8 Sample Size Based on BOR

| (45.1–69.2)<br>(47.6–71.5)<br>(50.1–73.8)<br>(52.7–76.0)<br>(55.2–78.2) |
|-------------------------------------------------------------------------|
| (50.1–73.8)<br>(52.7–76.0) |
| (52.7–76.0) |
| , |
| (55.2–78.2) |
| 95% CI (within the treatment group) [%] |
| (21.4–54.9) |
| (23.9–57.9) |
| (26.4–60.8) |
| (29.1–63.6) |
| (31.8–66.4) |

N (T-DM1 and capecitabine) / N (T-DM1) = 2

Expected BOR rate for patients who received trastuzumab emtansine of 43.6% (95% CI: 38.6%–48.6%) was chosen based on previously published data for T-DM1 in patients with unresectable, locally advanced or mBC previously treated with a taxane and trastuzumab (EMILIA study; Verma et al. 2012).

The BOR rates for patients treated with the combination of T-DM1 and capecitabine were chosen based on recent results from other combination studies of T-DM1 plus chemotherapy or trastuzumab plus capecitabine. Response rates were based on those observed in patients with HER2-positive mBC in a Phase Ib/IIa study (BP22752) that compared the combination of trastuzumab emtansine with docetaxel, with or without pertuzumab (ORR: 76% [95% CI: 53%–92%]), and also in a Phase II study that compared the combination of trastuzumab with docetaxel, with or without capecitabine (ORRs: 72.7% [95% CI: 63.4%–80.8%] and 70.5% [95% CI: 61.2%–78.8%]; Wardley et al., 2010).

Increased BOR rates for the combination treatment compared with single-agent trastuzumab emtansine are in line with previously published results of a randomized Phase III study in patients with locally advanced or mBC treated with the combination of trastuzumab with capecitabine *versus* capecitabine alone (ORR: 48.1% *versus* 27.0%, odds ratio = 2.50, p = 0.0115; von Minckwitz et al., 2009).

The precision for the BOR estimate of the combination of T-DM1 and capecitabine is approximately 12%, e.g. BOR of 60%, 95% CI of (47.6%, 71.5%). Due to the lower sample size of the treatment group T-DM1, the corresponding precision for the BOR estimate is increased to 18%, e.g. BOR of 46%, 95% CI of (29.1%, 63.6%).

The 2:1 randomization ratio will be applied to allow more patients being exposed to the combination of T-DM1 and capecitabine and to enable a more thorough assessment of the corresponding safety profile.

The estimation of sample size was performed by Nquery<sup>®</sup> and SAS<sup>®</sup> programs.

#### Stratification Factors

The following stratification factor will be implemented in the Randomized Phase II of the trial:

 Number of prior lines of treatment for metastatic disease (1 or >1; excluding single-agent hormones)

A treatment line is any regimen given to patient from treatment initiation until confirmed disease progression.

# Sample Size for Phase I: mGC

This part will be based on a classical 3 plus 3 Phase I design. From 3 to 12 patients might be enrolled into Cohort 2. There is no formal sample size estimation for this part.

# 6.2 SUMMARIES OF CONDUCT OF STUDY

# Phase I: Patients with mBC

Due to a small sample size, per-protocol (PP) population will not be defined for the Phase I, Cohort 1.

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 2, 03 September 2013

Major protocol violations will be summarized by treatment dosage. A median follow-up will be estimated for Phase I, Cohort 1.

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

For the Randomized Phase II part of the study, a PP population will be defined (Section 6.4).

Patient enrollment, duration of follow-up, discontinuation from study treatment and study, and reasons for discontinuation will be summarized by treatment group for all randomized patients. In addition, major protocol violations will be summarized by treatment arm.

# Phase I: Patients with mGC

Due to a small sample size, a PP population will not be defined for the Phase I. Cohort 2.

Major protocol violations will be summarized by treatment dosage. A median follow-up will be estimated for Phase I, Cohort 2.

# 6.3 SUMMARIES OF TREATMENT GROUP COMPARABILITY

#### Phase I: mBC

As Phase I is the Dose Finding part of the study, there are no treatment group comparisons for this part of the study.

Demographics, medical history, and baseline characteristics will be summarized. Continuous variables will be summarized by means of median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range while categorical variables – by the number and percentage of patients for each treatment dosage.

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

The Randomized Phase II part of the study is designed to explore the efficacy and safety of the combination of T-DM1 and capecitabine compared with T-DM1.

Demographics, medical history, and baseline characteristics will be summarized. Continuous variables will be summarized by means of median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range while categorical variables – by the number and percentage of patients for each treatment group.

# Phase I: mGC

As Phase I is the Dose Finding part of the study, there are no treatment group comparisons for this part of the study.

Demographics, medical history and baseline characteristics will be summarized. Continuous variables will be summarized by means of median,

# Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range while categorical variables – by the number and percentage for each treatment dosage.

# 6.4 EFFICACY ANALYSES

# Phase I, Cohort 1: mBC

The main analysis population will be the DLT evaluable population as defined in Section 6.5.

# Randomized Phase II: Exploration of Efficacy in mBC

The main analysis population for the efficacy analysis will be the intent-to-treat population (ITT), which will include all patients in the Randomized Phase II part of the study. The PP population will include all ITT patients who have at least one post-baseline tumor assessment during the Phase II and no major protocol violations, which will be defined in the statistical analysis plan (SAP).

# Phase I, Cohort 2: mGC

The main analysis population will be the DLT evaluable population as defined in Section 6.5.

#### 6.4.1 PRIMARY EFFICACY ENDPOINT

# Phase I, Cohort 1: Patients with mBC

The primary objectives are reaching the MTD and establishing a safety profile. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination.

ORR, as a main efficacy endpoint, will be assessed via BOR rate. The BOR is defined as the best response recorded from the date of enrollment until disease progression/recurrence, death, withdrawal of consent or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

# Randomized Phase II: Exploration of Efficacy in mBC

The primary efficacy endpoint for the Randomized Phase II part of the study is the ORR as assessed via BOR. The BOR is defined as the best response recorded from the start or randomization into the Phase II part of the study and until disease progression/recurrence, death, withdrawal of consent or EOS, whichever occurs first. To be assigned a status of PR or CR, i.e., to be a responder, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 28 days after the criteria for response are first met, i.e., patients need to have two consecutive assessments of PR or CR.

The emphasis of the exploratory Randomized Phase II part of the study will not be formal statistical hypothesis testing but the estimation of:

- The BOR rate with corresponding 95% CIs for each treatment group. The
  justification of the sample size is based on considerations regarding the
  width of 95% CIs for each treatment group estimate (precision of the
  corresponding estimate).
- The treatment effect (between treatment groups comparison) with corresponding 95% CIs.

The number and proportions of responders and non-responders (based on BOR) together with 95% Clopper-Pearson Cls will be presented for each treatment group.

The difference in BOR between treatment groups will be displayed with associated 95% CIs using the Hauck-Anderson approach.

Logistic analysis will be used to assess the influence of the stratification factor and baseline covariates in an exploratory manner.

# Phase I, Cohort 2: Patients with mGC

The primary objectives are reaching the MTD and establishing a safety profile. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination.

ORR, as a main efficacy endpoint, will be assessed via BOR rate. The BOR is defined as the best response recorded from the date of enrollment until disease progression/recurrence, death, withdrawal of consent or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

# 6.4.2 SECONDARY EFFICACY ENDPOINTS

# Phase I, Cohort 1: mBC

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

# Randomized Phase II: Exploration of Efficacy in mBC

The secondary efficacy endpoints for the Randomized Phase II will be:

- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

TTR is defined as the time from randomization to first documentation of confirmed PR or CR (whichever occurs first). Patients who do not have a confirmed response will be censored at the date of the last tumor assessment.

DoR is defined as the period from the date of initial confirmed PR or CR until the date of PD or death from any cause. Patients with no documented progression after CR or PR will be censored at the last date, at which they are known to have had the CR or PR, respectively. The method for handling censoring is the same as described for the PFS below. Only patients with BOR of CR or PR (i.e., responders) will be included in the analysis of DoR.

For patients with a BOR of CR or PR, TTR is defined as the time from randomization to the date of first CR or PR. The censoring rules will be similar to those of the PFS.

TTP is defined as time from randomization to the first occurrence of PD. Patients who have not progressed at the time of study completion (including patients who have died before PD) or who are lost to follow-up are censored at the date of the last tumor assessment.

TTF is defined as time from randomization until treatment failure, e.g., to disease progression, death, withdrawal due to AE or laboratory abnormality, or refusal of treatment. Patients who do not experience any of the above events while on study will be censored on the day of their last tumor assessment.

PFS is defined as time from randomization until the first documented progression of disease or death from any cause, whichever occurs first. Patients with no PFS events will be censored at the time of the last evaluable tumor assessment. Patients with no tumor assessment after the baseline visit at the time of Phase II will be censored at the time of enrollment plus 1 day. OS is defined as the time from randomization until the date of death, regardless of the cause of death. Patients who were alive at the time of the analysis will be censored at the date of the last follow-up assessment.

Estimates for the survivor function of both treatment groups for TTR, DoR, TTP, TTF, and OS will be obtained by using the Kaplan-Meier method. HRs and associated 95% CIs will be estimated from non-stratified and stratified (based on the stratification factor) Cox regression models.

Clinical benefit response includes patients whose best (confirmed) response was PR, CR or SD that lasted at least 6 months. CBR will be summarized in a similar way to the primary efficacy endpoint, ORR as assessed by BOR.

# Phase I, Cohort 2: mGC

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

# 6.5 SAFETY ANALYSES

# Safety Population Phase I, Cohort 1: mBC

The DLT evaluable population is defined for all enrolled and treated patients who have not experienced any major protocol violation (including violation of the inclusion and exclusion criteria) and completed Cycle 1.

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

The safety population (SP) will include all patients who received at least one dose of study medication during Phase I. Safety endpoints will be summarized by treatment dosage.

Safety parameters will be analyzed in a similar way to safety parameters in Phase I, Cohort 2: mGC.

# Randomized Phase II: Exploration of Safety in mBC

The SP will include all patients who received at least one dose of study medication during the Randomized Phase II part of the study. Safety endpoints will be summarized by treatment group.

Safety endpoints during Phase II will be assessed via total AEs, AEs Grade ≥ 3, SAEs, AESIs (as described in Section 5), premature withdrawal from study medication, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by the Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Based on the safety profile of trastuzumab emtansine time to onset of the first episode of any AESI described in Section 5 will also be summarized via Kaplan-Meier estimates. Additional summaries by frequency tables will also be provided for the AESIs. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry will be presented in shift tables of NCI-CTC grade at baseline *versus* worst grade during treatment for the Randomized Phase II part of the study.

LVEF will be summarized over time by means of mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations, will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

# Safety Population Phase I, Cohort 2: mGC

The DLT evaluable population is defined for all enrolled and treated patients who have not experienced any major protocol violation (including violation of the inclusion and exclusion criteria) and have completed Cycle 1.

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

The SP will include all patients who received at least one dose of study medication during Phase I. Safety endpoints will be summarized by treatment dosage.

Safety parameters for this part of the study will be summarized by treatment dose. The summaries of AEs, SAEs, AEs that caused discontinuation from the study treatment, and AESIs will be analyzed in a similar way to AEs in Phase II.

The incidence of AEs and SAEs will be summarized according to the primary SOC and, within each SOC, by MedDRA preferred term. Based on the safety profile of trastuzumab emtansine time to onset of the first episode of any AESI described in Section 5 will also be summarized via Kaplan-Meier estimates. Additional summaries by frequency tables will also be provided for the AESIs. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry will be presented in shift tables of NCI-CTC grade at baseline versus worst grade during treatment for Phase I, Cohort 2, and overall.

LVEF will be summarized over time by means of mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### 6.6 PHARMACODYNAMIC ANALYSES

No pharmacodynamic analyses are planned for this study.

#### 6.7 PHARMACOKINETIC ANALYSES

# For Phase I only (Patients with mBC and mGC):

The following PK parameters of trastuzumab emtansine and capecitabine (including but not limited to those listed below) will be determined only in the Phase I part of the study for Cohort 1 and Cohort 2 in all patients who receive study treatment using either non-compartmental and/or population methods, if data allow:

Serum concentrations of trastuzumab emtansine (conjugate) and total trastuzumab

- Plasma concentrations of DM1, capecitabine and its active metabolite 5-FU
- Total exposure (e.g., AUC)
- C<sub>max</sub>
- Clearance (CL)
- V<sub>d</sub>
- T<sub>1/2</sub>

The PK of trastuzumab emtansine, total trastuzumab and DM1 will be compared with historical single-agent PK data to evaluate the potential effect of capecitabine on the PK of trastuzumab emtansine and related analytes. The PK of capecitabine and its active metabolite 5-FU in Cycle 1 (in the absence of trastuzumab emtansine) will be compared with the PK of Cycle 2 (in the presence of trastuzumab emtansine) to evaluate the potential effect of trastuzumab emtansine on the PK of capecitabine and 5-FU.

All PK parameters will be listed and tabulated by treatment dose and by Cohort. Descriptive summary statistics including arithmetic mean, geometric mean (e.g., AUC and  $C_{max}$ ), median, range, s.d., and coefficient of variation will be presented for each cohort. Nonlinear mixed effects modeling will be also used but details will be presented in the SAP.

PK samples can be obtained ad hoc in case of SAE or unexpected toxicities which may suggest a potential drug-drug interaction.

# 6.8 EXPLORATORY ANALYSES

For all patients a retrospective central confirmation of the HER2 status will be done. Further exploratory analysis for HER2-positive patients— (based on central confirmation) will be done for selected endpoints such as BOR and safety endpoints (AEs, SAEs, AEs with Grade ≥ 3 and AESIs).

# For the Randomized Phase II: Exploration of Efficacy and Safety in Patients with mBC only:

Subgroup analysis for BOR, safety endpoints (AEs, SAEs, AEs with Grade ≥ 3 and AESIs) in Phase II will be presented for: elderly *versus* younger patients, and patients with ECOG 0–1 *versus* ECOG 2.

More details about subgroups will be provided in the SAP.

# **Pharmacoeconomic Endpoint:**

The resource expenditure due to hospitalizations that are not study-defined evaluations while on study treatment will be evaluated. The number of hospital visits, number of days admitted, and type of visits (emergency department *versus* inpatient care) will be collected. The reason for admission (disease progression *versus* AE) will also be assessed.

# 6.9 INTERIM ANALYSES

There is no formal efficacy interim analysis. **Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd**Protocol MO28230, Version 2, 03 September 2013

However, an IDMC will advise whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 20 and 60 patients have received at least 3 cycles (Cycle 3 Day 1) of treatment in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the course of the Randomized Phase II of the study or as requested.

Efficacy data will only be provided if required by the IDMC to estimate the riskbenefit balance for the patients. Further details on the function and logistics of the IDMC will be provided in the IDMC Charter.

The design of this study includes: Phase I, Randomized Phase II and different cohorts. Corresponding analyses as described in the protocol will be performed when all data for particular cohort and study phase are collected and cleaned.

#### 7. DATA COLLECTION AND MANAGEMENT

#### 7.1 **DATA QUALITY ASSURANCE**

The Sponsor will be responsible for data management of this study, including quality checking of the data. Data entered manually will be collected via EDC using eCRFs. The sites will be responsible for data entry into the EDC system. In the event of discrepant data, the Sponsor will request data clarification from the sites, which the sites will resolve electronically in the EDC system.

The Sponsor will produce an EDC Study Specification document that describes the quality checking to be performed on the data. Central laboratory data and other electronic data will be sent directly to the Sponsor, using the Sponsor's standard procedures to handle and process the electronic transfer of these data.

eCRFs and correction documentation will be maintained in the EDC system's audit trail. System backups for data stored by the Sponsor and records retention for the study data will be consistent with the Sponsor's standard procedures.

#### 7.2 **ELECTRONIC CASE REPORT FORMS**

eCRFs are to be completed using a Sponsor-designated EDC system. Sites will receive training and have access to a manual for appropriate eCRF completion. eCRFs will be submitted electronically to the Sponsor and should be handled in accordance with instructions from the Sponsor.

All eCRFs should be completed by designated, trained site staff. eCRFs should be reviewed and electronically signed and dated by the investigator or a designee.

At the end of the study, the investigator will receive patient data for his or her site in a readable format on a compact disc that must be kept with the study records. Acknowledgment of receipt of the compact disc is required.

# 7.3 SOURCE DATA DOCUMENTATION

Study monitors will perform ongoing SDV to confirm that critical protocol data (i.e., source data) entered into the eCRFs by authorized site personnel are accurate, complete, and verifiable from source documents.

Source documents (paper or electronic) are those in which patient data are recorded and documented for the first time. They include, but are not limited to, hospital records, clinical and office charts, laboratory notes, memoranda, patient-reported outcomes, evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies of transcriptions that are certified after verification as being accurate and complete, microfiche, photographic negatives, microfilm or magnetic media, X-rays, patient files, and records kept at pharmacies, laboratories, and medico-technical departments involved in a clinical trial.

Source documents that are required to verify the validity and completeness of data entered into the eCRFs must not be obliterated or destroyed.

To facilitate SDV, the investigators and institutions must provide the Sponsor with direct access to applicable source documents and reports for trial-related monitoring, Sponsor audits, and IRB/EC review. The investigational site must also allow inspection by applicable health authorities.

# 7.4 USE OF COMPUTERIZED SYSTEMS

When clinical observations are entered directly into an investigational site's computerized medical record system (i.e., in lieu of original hardcopy records), the electronic record can serve as the source document if the system has been validated in accordance with health authority requirements pertaining to computerized systems used in clinical research. An acceptable computerized data collection system (for clinical research purposes) would be one that (1) allows data entry only by authorized individuals; (2) prevents the deletion or alteration of previously entered data and provides an audit trail for such data changes (e.g., modification of file); (3) protects the database from tampering; and (4) ensures data preservation.

In collaboration with the study monitor, Sponsor's Quality Assurance group may assist in assessing whether electronic records generated from computerized medical record systems used at investigational sites can serve as source documents for the purposes of this protocol.

If a site's computerized medical record system is not adequately validated for the purposes of clinical research (as opposed to general clinical practice), applicable hardcopy source documents must be maintained to ensure that critical protocol data entered into the eCRFs can be verified.

# 7.5 RETENTION OF RECORDS

U.S. FDA regulations (21 Code of Federal Regulations §312.62[c]) and the ICH Guideline for Good Clinical Practice (GCP) (see Section 4.9 of the guideline) require that records and documents pertaining to the conduct of this study and the distribution of investigational drug, including eCRFs, Consent


Forms, laboratory test results, and medication inventory records, must be retained by the Principal Investigator for 2 years after the last marketing application approval in an ICH region or after at least 2 years have elapsed since formal discontinuation of clinical development of the investigational product. All state and local laws for retention of records also apply.

No records should be disposed of without the written approval of the Sponsor. Written notification should be provided to the Sponsor for transfer of any records to another party or moving them to another location.

For studies conducted outside the United States under a U.S. Investigational New Drug (IND) application, the Principal Investigator must comply with the record retention requirements set forth in the U.S. FDA IND regulations and the relevant national and local health authorities, whichever is longer.

# 8. <u>ETHICAL CONSIDERATIONS</u>

# 8.1 COMPLIANCE WITH LAWS AND REGULATIONS

This study will be conducted in full conformance with the ICH E6 guideline for GCP and the principles of the Declaration of Helsinki, or the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual. The study will comply with the requirements of the ICH E2A guideline (Clinical Safety Data Management: Definitions and Standards for Expedited Reporting). Studies conducted in the United States or under a U.S. IND application will comply with U.S. FDA regulations and applicable local, state, and federal laws. Studies conducted in the European Union (EU)/European economic area (EEA) will comply with the EU Clinical Trial Directive (2001/20/EC).

# 8.2 INFORMED CONSENT

Sponsor's Sample Informed Consent Form will be provided to each site. If applicable, it will be provided in a certified translation of the local language. The Sponsor or its designee must review and approve any proposed deviations from the Sample Informed Consent Form or any alternate Consent Forms proposed by the site before IRB/EC submission. The final IRB/EC-approved Consent Forms must be provided to the Sponsor for health authority submission purposes according to local requirements.

The Consent Form must be signed and dated by the patient or the patient's legally authorized representative before his or her participation in the study. The case history or clinical records for each patient shall document the informed consent process and that written informed consent was obtained prior to participation in the study.

A copy of each signed Consent Form must be provided to the patient or the patient's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

All signed and dated Consent Forms must remain in each patient's study file and must be available for verification by study monitors at any time.

The Informed Consent Form should be revised whenever there are changes to procedures outlined in the informed consent or when new information becomes available that may affect the willingness of the patient to participate.

For any updated or revised Consent Forms, the case history for each patient shall document the informed consent process and that written informed consent was obtained for the updated/revised Consent Form for continued participation in the study. The final revised IRB/EC-approved Informed Consent Form must be provided to the Sponsor for regulatory purposes.

If the site uses a separate Authorization Form for patient authorization to use and disclose personal health information under the U.S. Health Insurance Portability and Accountability Act (HIPAA) regulations, the review, approval, and other processes outlined above apply except that IRB/IEC review and approval may not be required per study site policies.

# 8.3 INSTITUTIONAL REVIEW BOARD OR ETHICS COMMITTEE

This protocol, the Informed Consent Forms, any information to be given to the patient, and relevant supporting information must be submitted to the IRB/EC by the Principal Investigator and reviewed and approved by the IRB/EC before the study is initiated. In addition, any patient enrollment materials must be approved by the IRB/EC.

The Principal Investigator is responsible for providing written summaries of the status of the study to the IRB/EC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC. Investigators are also responsible for promptly informing the IRB/EC of any protocol amendments.

In addition to the requirements to report protocol-defined AEs to the Sponsor, investigators are required to promptly report to their respective IRB/EC all unanticipated problems involving risk to human patients. Some IRBs/ECs may want prompt notification of all SAEs, whereas others require notification only about events that are serious, assessed to be related to study treatment, and are unexpected. Investigators may receive written IND safety reports or other safety related communications from the Sponsor. Investigators are responsible for ensuring that such reports are reviewed and processed in accordance with regulatory requirements and with the policies and procedures established by their IRB/EC and archived in the site's study file.

# 8.4 CONFIDENTIALITY

The Sponsor maintains confidentiality standards by coding each patient enrolled in the study through assignment of a unique patient identification number. This means that patient names are not included in data sets that are transmitted to any Sponsor location.

Patient medical information obtained by this study is confidential and may only be disclosed to third parties as permitted by the Informed Consent Form (or separate authorization for use and disclosure of personal health information) signed by the patient, unless permitted or required by law.

Medical information may be given to a patient's personal physician or other appropriate medical personnel responsible for the patient's welfare, for treatment purposes.

Data generated by this study must be available for inspection upon request by representatives of the U.S. FDA and other national and local health authorities, the Sponsor monitors, representatives, and collaborators, and the IRB/EC for each study site, as appropriate.

# 8.5 FINANCIAL DISCLOSURE

Investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate health authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

# 9. <u>STUDY DOCUMENTATION, MONITORING, AND ADMINISTRATION</u>

# 9.1 STUDY DOCUMENTATION

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented, including but not limited to the protocol, protocol amendments, Informed Consent Forms, and documentation of IRB/EC and governmental approval. In addition, at the end of the study, the investigator will receive the patient data, which includes an audit trail containing a complete record of all changes to data.

# 9.2 SITE INSPECTIONS

Site visits will be conducted by the Sponsor or an authorized representative for inspection of study data, patients' medical records, and eCRFs. The investigator will permit national and local health authorities, the Sponsor monitors, representatives, and collaborators, and the IRBs/ECs to inspect facilities and records relevant to this study.

# 9.3 ADMINISTRATIVE STRUCTURE

The study will have a SC, iDMC, central laboratory, IxRS, eCRF, and will be conducted by a contract research organization (CRO) together with the Sponsor.

# 9.4 PUBLICATION OF DATA AND PROTECTION OF TRADE SECRETS

The results of this study may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or

Study MO28230

abstracts to the Sponsor prior to submission. This allows the Sponsor to protect proprietary information and to provide comments based on information from other studies that may not yet be available to the investigator.

The Sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter trials only in their entirety and not as individual center data. In this case, a coordinating investigator will be designated by mutual agreement.

Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements. Any formal publication of the study in which contribution the Sponsor personnel exceeded that of conventional monitoring will be considered as a joint publication by the investigator and the appropriate the Sponsor personnel.

Any inventions and resulting patents, improvements, and/or know-how originating from the use of data from this study will become and remain the exclusive and unburdened property of the Sponsor, except where agreed otherwise.

# 9.5 PROTOCOL AMENDMENTS

Any protocol amendments will be prepared by the Sponsor. Protocol amendments will be submitted to the IRB/EC and to regulatory authorities in accordance with local regulatory requirements.

Approval must be obtained from the IRB/EC and regulatory authorities (as locally required) before implementation of any changes, except for changes necessary to eliminate an immediate hazard to patients or changes that involve logistical or administrative aspects only (e.g., change in Medical Monitor or contact information).

# 10. REFERENCES

- 1. Albarello L, Pecciarini L, Doglioni C. HER2 testing in gastric cancer. Adv Anat Pathol 2011; 18:53–9.
- 2. Austin CD, De Mazière AM, Pisacane PI, et al. Endocytosis and sorting of ErbB2 and the site of action of cancer therapeutics trastuzumab and geldanamycin. Mol Biol Cell 2004; 15:5268–82.
- Bang YJ, van Cutsem E, Feyereislova A, et al. Trastuzumab in combination with chemotherapy *versus* chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet 2010; 376:687–97.
- 4. Blum JL, Dieras V, Lo Russo PM, et al. Multicenter, Phase II study of oral capecitabine in taxane-pretreated metastatic breast carcinoma patients. Cancer 2001; 92:1759–68.
- 5. Blum JL, Jones SE, Buzdar AU, et al. Multicenter Phase II study of capecitabine in paclitaxel-refractory metastatic breast cancer. J Clin Oncol 1999; 17:485–93.
- 6. Cabanillas F, Chan KK, Floss HG, et al. Results of a Phase II study of maytansine in patients with breast carcinoma and melanoma. Cancer Treat Rep 1979; 63:507–9.
- 7. Cassady JM, Chan KK, Floss HG, et al. Recent developments in the maytansinoid antitumor agents. Chem Pharm Bull (Tokyo) 2004; 52:1–26.
- 8. Catalano V, Labianca R, Beretta GD, et al. Gastric cancer. Crit Rev Oncol Hematol 2005; 54:209–41.
- 9. Igawa Y, Matsubara M, Matsunaga K, et al. Pharmacokinetic (PK) and pharmacodynamic (PD) analysis of trastuzumab emtansine (T-DM1) in Japanese patients with advanced or recurrent HER2-positive breast cancer (JO22591): Comparison with Western patients. ASCPT 2012.
- 10. De Vivo R, Pignata S, Palaia R, et al. The role of chemotherapy in the management of gastric cancer. J Clin Gastroenterol 2000; 30:364–71.
- 11. Erickson HK, Park PU, Widdison WC, et al. Antibody-maytansinoid conjugates are activated in targeted cancer cells by lysosomal degradation and linker-dependent intracellular processing. Cancer Res 2006; 66:4426–33.
- 12. Faivre J, Forman D, Esteve J, et al. Survival of patients with oesophageal and gastric cancers in Europe. Eur J Cancer 1998; 34:2167–75.
- 13. Ferlay J, Shin HR, Bray F, et al. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer 2010; 127:2893–917.
- 14. Geyer CE, Forster J, Lindquist D, et al. Lapatinib plus capecitabine for HER2-positive advanced breast cancer. N Engl J Med 2006; 355:2733–43.
- 15. Girish S, Gupta M, Wang B, et al. Clinical pharmacology of trastuzumab emtansine (T-DM1): an antibody–drug conjugate in development for the

- treatment of HER2-positive cancer. Cancer Chemother Pharmacol 2012; 69:1229–40.
- 16. Gupta M, LoRusso PM, Wang B, et al. Clinical implications of pathophysiological and demographic covariates on the population pharmacokinetics of trastuzumab-DM1, a HER2-targeted antibody–drug conjugate, in patients with HER2-positive metastatic breast cancer. J Clin Pharmacol 2011; 52:691–703.
- 17. Hofmann M, Stoss O, Shi D, et al. Assessment of a HER2 scoring system for gastric cancer: results from a validation study. Histopathology 2008; 52:797–805.
- 18. Issell BF, Crooke ST. Maytansine. Cancer Treat Rev 1978; 5:199–207.
- 19. Jemal A, Bray F, Center MM, et al. Global Cancer Statistics. CA Cancer J Clin 2011; 61:69–90.
- 20. Junttila TT, Li G, Parsons K, et al. Trastuzumab-DM1 (T-DM1) retains all the mechanisms of action of trastuzumab and efficiently inhibits growth of lapatinib insensitive breast cancer. Breast Cancer Res Treat 2011; 128:347–56.
- 21. Krop IE, Beeram M, Modi S, et al. Phase I study of trastuzumab-DM1, an HER2 antibody-drug conjugate, given every three weeks to patients with HER2-positive metastatic breast cancer. J. Clin Oncol 2010; 28:2698–704.
- 22. Krop IE, Mita M, Burris HA, et al. A Phase I Study of Weekly Dosing of Trastuzumab-DM1 (T-DM1) in Patients with Advanced HER 2-Positive Breast Cancer. Clin Oncol 2008; 26 (Suppl):abstract1029.
- 23. Krop IE, Mita M, Burris HA, et al. A Phase I study of weekly dosing of trastuzumab-DM1 (T-DM1) in patients with advanced HER2+ breast cancer. (SABCS 2008) Cancer Res 2009; 69 (Suppl 1):3136.
- 24. Lewis Phillips G, Fields CT, Crocker L, et al. Potent anti-tumor activity of trastuzumab-DM1 antibody conjugate in combination with cytotoxic chemotherapeutic agents, antibodies or small molecule kinase inhibitors. AACR 2008; poster#2133.
- 25. Marty M, Cognetti F, Maraninchi D, et al. Randomized Phase II trial of the efficacy and safety of trastuzumab combined with docetaxel in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer administered as first-line treatment: the M77001 study group. J Clin Oncol 2005; 23:4265–74.
- 26. Moldoveanu Z, Huang W-Q, Kulhavy R, et al. Human male genital tract secretions: both mucosal and systemic immune compartments contribute to the humoral immunity. J Immunol 2005; 175:4127–36.
- 27. Parkin DM, Bray F, Ferlay J, et al. Global Cancer Statistics 2002. CA Cancer J Clin. 2005; 55:74–108.
- 28. Power DG, Kelsen DP, Shah MA. Power Advanced gastric cancer--slow but steady progress. Cancer Treat Rev 2010; 36:384-92.
- 29. Press MF, Sauter G, Bernstein L, et al. Diagnostic evaluation of HER-2 as a molecular target: an assessment of accuracy and reproducibility of

- laboratory testing in large, prospective, randomized clinical trials. Clin Cancer Res 2005; 11:6598–607.
- 30. Ries LAG, Melbert D, Krapcho M, et al (eds). SEER Cancer Statistics Review 1975 2005. Bethesda (MD): National Cancer Institute, 2008;http://seer.cancer.gov/csr/1975\_2005
- 31. Sawaki A, Ohashi Y, Omuro Y, et al. Efficacy of trastuzumab in Japanese patients with HER2-positive advanced gastric or gastroesophageal junction cancer: a subgroup analysis of the Trastuzumab for Gastric Cancer (ToGA) study. Gastric Cancer 2012; 15:313–22.
- 32. Shen B-Q, Bumbaca D, Saad O, et al. Metabolic Fate and Pharmacokinetic Characterization of Trastuzumab Emtansine (T-DM1): An Emphasis on Preclinical and Clinical Catabolism. ASCPT 2011.
- 33. Slamon DJ, Clark GM, Wong SG, et al. Human breast cancer; correlation of relapse and survival with amplification of the HER2/neo oncogene. Science 1987; 235:177–82.
- 34. Slamon DJ, Leyland-Jones B, Shak S, et al. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med 2001; 344:783–92.
- 35. Spector NL, Xia W, Burris H 3<sup>rd</sup>, et al. Study of the biologic effects of lapatinib, a reversible inhibitor of ErbB1 and ErbB2 tyrosine kinases, on tumor growth and survival pathways in patients with advanced malignancies. J Clin Oncol 2005; 23:2502–12.
- 36. Sundaresan S, Penuel E, Sliwkowski MX. The biology of human epidermal growth factor receptor 2. Curr Oncol Rep 1999; 1:16–22.
- 37. Tanner M, Hollmen M, Junttila TT, et al. Amplification of HER2 in gastric cancer—association with topoisomerase IIa gene amplification, intestinal type, poor prognosis and sensitivity to trastuzumab. Ann Oncol 2005; 16:273–8.
- 38. Therasse P, Eisenhauer EA, Verwij J. RECIST revisited: a review of validation studies on tumour assessment. Eur J Cancer 2000; 42:1031–9.
- 39. Tjulandin S, Makhson A, Gligorov J, et al. First results of a Phase II study of Bevacizumab in combination with trastuzumab and capecitabine as first-line treatment of HER2-positive LR/MBC. ASCO 2011; Poster #571.
- 40. Verma S, Miles D, Gianni L, et al. Trastuzumab emtansine for HER2-positive advanced breast cancer. N Engl J Med 2012; 367:1783–91.
- 41. von Minckwitz G, Schwedler K, Schmidt M, et al. Trastuzumab beyond progression: overall survival analysis of the GBG 26/BIG 3-05 Phase III study in HER2-positive breast cancer. Eur J Cancer 2011; 47:2273–81.
- 42. Yang J, Wang Y, Zhao H, et al. Combination of exposure-response and case-control analyses in regulatory decision making. J Clin Oncol 2011; 29: (Suppl); 4087.
- 43. Yoon HH, Shi Q, Sukov WR, et al. Association of HER2/ErbB2 expression and gene amplification with pathologic features and prognosis in esophageal adenocarcinomas. Clin Cancer Res 2012; 18:546–54.
Trastuzumab Emtansine 301 RO5304020 Study MO28230

44. Wardley A, Anton-Torres A, Pivot X, et al. Trastuzumab plus docetaxel with or without capecitabine in patients with HER2-positive advanced/metastatic breast cancer: first efficacy results from the Phase II MO16419 (CHAT) Study. SABCS 2006; Abstract# 2063.

- 45. Wardley A, Pivot X, Morales-Vasquez F, et al. Randomized phase II trial of first-line trastuzumab plus docetaxel and capecitabine compared with trastuzumab plus docetaxel in HER2-positive metastatic breast cancer. J Clin Oncol. 2010; 28:976-83.
- 46. World Health Organization, World Health Statistics 2011; http://www.who.int/whosis/whostat/2011/en/

Kadcyla (RO5304020) Roche Clinical Study Report - Protocol MO28230

### Appendix 1 Schedule of Assessments

Table 1 Schedule of assessments for mBC patients (Phase I, Cohort 1 and Randomized Phase II)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | | Сус | cle 4 Onwa | ards | Safety<br>Follow-Up<br>Visit | Follow-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 3-6<br>months |
| Informed Consent | X <sup>a</sup> | | | | | | | | | | | |
| HER2 Status | Xp | | | | | | | | | | | |
| Medical History and Demographics | Х | | | | | | | | | | | |
| Complete Physical Examination | Х | | | | | | | | | | | |
| Limited Physical Examination <sup>c</sup> | | Х | | | Х | | | Х | | | Х | |
| Height and Weight <sup>d</sup> | Х | Х | | | Х | | | Х | | | Х | |
| Vital Signs <sup>e</sup> | Х | Х | | | Х | | | Х | | | Х | |
| ECOG Performance Status | Х | Х | | | Х | | | Х | | | Х | |
| Concomitant Medication Reporting | X <sup>f</sup> | Х | | | | | Ongoir | ng | | | | |
| AE Reporting | X <sup>g</sup> | | • | | | Ongoing | | | | | Х | X <sup>h</sup> |
| 12-lead ECG | Х | | | | | | | | | | | |
| ECHO/MUGA <sup>i</sup> | X <sup>i</sup> | | | Xi | | | X <sup>i</sup> | | | X <sup>i</sup> | X <sup>i</sup> | |
| Tumor Assessments <sup>j</sup> | Х | | | ks after rar | r early dis | | on, until di | | | | х | х |
| Brain CT or MRI <sup>k</sup> | Х | | ı | At the disc | retion of th | ne investig | ator, if clin | ically indi | cated, unti | l disease p | rogression | |
| Bone Scan/Imaging <sup>I</sup> | Х | | | | | , | As clinicall | y indicate | d | | | |

### Table 1Schedule of assessments for mBC patients (Phase I, Cohort 1 and Randomized Phase II) (cont.)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | Cyc | le 4 Onwa | rds | Safety<br>Follow-Up<br>Visit | Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 3-6<br>months |
| Hematology <sup>m</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | | | Х | |
| Biochemistry <sup>o</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | | | Х | |
| Urinalysis <sup>p</sup> | Х | | | | As clin | ically indic | ated | | | | Х | |
| INR/aPTT | Х | As clinically indicated, e.g. for patients receiving anticoagulation therapy | | | | | Х | | | | | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Χ <sup>q</sup> | | | Χ <sup>q</sup> | Х | Х |
| PK/PD Samples (see Appendix 2) <sup>r</sup> | | X <sup>r</sup> | | | X <sup>r</sup> | | | | | | | |
| Assessment of Patient<br>Hospitalizations and/or Hospital<br>Visits | | х | | | Х | | | х | | | х | |
| Administration of Trastuzumab Emtansine | | D 2 <sup>s</sup> | | | D 1 <sup>s</sup> | | | D 1 <sup>s</sup> | | | | |
| Administration of Capecitabine | | D · | 1–14 | | D 1 | -14 | | D 1 | -14 | | | |
| Overall Survival | Х | | | | | Х | | | | | Х | Х |
| Randomization into the Phase II Part of the Study | X <sup>t</sup> | | | | | | | | | | | |

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

- 1.NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within **14 days** prior to first treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1).
- 2.All patients will be followed-up every 6 months (except for pregnancy, which is at 3 and 6 months after safety follow-up visit until disease progresses for tumor assessment or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than disease progression will continue to undergo tumor assessments every 3–6 months.
- a)Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests.
- b)HER2-positivity is defined as IHC 3+ or gene amplification by ISH. It will be performed locally for patients with mBC.
- c)Limited symptom-directed physical examination.
- d)Height to be obtained at screening or at Cycle 1 Day 1 only.
- e)Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f)Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to first study treatment.
- g)During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h)Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatment-related AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i)Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, and on Day 15-21 of Cycle 1, Cycle 3 and every third cycle thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

- j)Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than PD, continued tumor assessments according to the protocol every 3–6 months.
- k)Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 4 months) as detailed in Section 4.5.1.4 of the protocol and in Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- I)An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- m)Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and white blood cells (WBC) with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils.
- n)Assessments should be performed at screening, on Day 1, 8 and 15 of Cycles 1–3, on Day 1 of all subsequent cycles, and weekly following any hematologic AE. If capecitabine is discontinued due to toxicity, assessments should be performed weekly (minimum) until resolution of the AE (Grade ≤ 1/ baseline), and on Day 1 of subsequent cycles thereafter. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- o)Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, blood urea nitrogen (BUN), creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN).
- p)Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.

- q)Serum β-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.
- r)Pharmacokinetic assessments will be performed during the Dose Finding part of the study only (see Appendix 2).
- s)Trastuzumab emtansine will be administered on Day 1 of each 3-weekly cycle for all patients with mBC in Cohort 1 and Randomized Phase II period of the study except in the first cycle where trastuzumab emtansine will be given on Day 2 (to allow PK sampling).
- t)Patients will be randomized only in the Randomized Phase II part of the study. No blinding will be used, as this is an open-label study. A 2:1 randomization ratio will be applied to allow more patients to be exposed to the combination of T-DM1 and capecitabine, and to enable a more thorough assessment of the corresponding safety profile.

Kadcyla (RO5304020) Roche Clinical Study Report - Protocol MO28230

### Appendix 1 Schedule of Assessments (cont.)

### Table 2 Schedule of assessments for patients with mGC (Phase I, Cohort 2)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2-3 | 3 | Сус | cle 4 Onw | ards | Safety<br>Follow-Up<br>Visit | Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28–42 days<br>after last<br>dose | every 3–6<br>months |
| Informed Consent | X <sup>a</sup> | | | | | | | | | | | |
| HER2 Status | Xp | | | | | | | | | | | |
| Medical History and Demographics | Х | | | | | | | | | | | |
| Complete Physical Examination | Х | | | | | | | | | | | |
| Limited Physical Examination <sup>c</sup> | | Х | | | Х | | | Х | | | Х | |
| Height and Weight <sup>d</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Vital Signs <sup>e</sup> | Х | Х | | | Х | | | Х | | | Х | |
| ECOG Performance Status | Х | Х | | | Х | | | Х | | | Х | |
| Concomitant Medication Reporting | X <sup>f</sup> | Х | | | | | Ongoi | ng | | | | |
| AE Reporting | X <sup>g</sup> | | | | | Ongoing | | | | | Х | X <sup>h</sup> |
| 12-lead ECG | Х | | | | | | | | | | | |
| ECHO/MUGA <sup>i</sup> | X <sup>i</sup> | | | X <sup>i</sup> | | | Xi | | | X <sup>i</sup> | X <sup>i</sup> | |
| Tumor Assessments <sup>j</sup> | х | At 9 weeks after C1D1, and every 12 weeks thereafter, regardless of dose delay or early discontinuation, until disease progression or study termination | | | | Х | | | | | | |
| Brain CT or MRI <sup>k</sup> | Х | | | At the disc | cretion of | the investig | ator, if clir | nically indic | cated, until | l disease p | rogression | • |
| Bone Scan/Imaging <sup>l</sup> | Х | | | | | | As clinical | ly indicate | d | | | |

### Table 2 Schedule of assessments for patients with mGC (Phase I, Cohort 2) (cont.)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2- | -3 | Су | cle 4 Onv | vards | Safety<br>Follow-Up<br>Visit | Follow-Up <sup>3</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28–42 days<br>after last<br>dose | every 3–6<br>months |
| Hematology <sup>m</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | Х | |
| Biochemistry <sup>o</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | Х | |
| Urinalysis <sup>p</sup> | Х | | | | As c | linically in | dicated | | | | Х | |
| INR/aPTT | Х | P | As clinically indicated, e.g. for patients receiving anticoagulation therapy | | | | | Х | | | | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Xq | | | X <sup>q</sup> | Х | Х |
| PK/PD Samples (see Appendix 2) | | Х | | | Х | | | | | | | |
| Assessment of Patient<br>Hospitalizations and/or Hospital<br>Visits | | х | | | Х | | | Х | | | Х | |
| Administration of Trastuzumab Emtansine | | D 2 <sup>r</sup> | Х | х | Х | Х | Х | Х | х | Х | | |
| Administration of Capecitabine | | D 1- | -14 | | D 1 | -14 | | D 1 | -14 | | | |
| Overall Survival | Х | | | • | • | Х | | | | | Х | Х |

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

- 1.NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within **14 days** prior to first study treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1) visit.
- 2.All patients will be followed-up every 6 months (except for pregnancy, which is at 3 and 6 months after safety follow-up visit) until disease progresses for tumor assessment or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than disease progression will continue to undergo tumor assessments every 3–6 months.
- a)Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests.
- b)HER2-positivity is defined as IHC 3+ alone or IHC 2+ in combination with gene amplification by ISH. For patients with mGC enrolled into Cohort 2, central confirmation of HER2 status is required.
- c)Limited symptom-directed physical examination.
- d)Height to be obtained at screening or at Cycle 1 Day 1 only.
- e)Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f)Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to fist study treatment.
- g)During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h)Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatment-related AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i)Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, and on Days 15–21, 30–42 and 9 weeks thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

- j)Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than PD, continued tumor assessments according to the protocol every 3–6 months.
- k)Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 4 months) as detailed in Section 4.5.1.4 of the protocol and in Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- I)An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to first study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- m)Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and WBC with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils).
- n)Assessments should be performed at screening, on Day 1, 8 and 15 of all cycles. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- o)Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, BUN/urea, creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN).
- p)Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.
- q)Serum β-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.
- r)Trastuzumab emtansine will be administered on Day 1 of each weekly cycle for all patients enrolled in Cohort 2 (A&B) except in the first cycle where trastuzumab emtansine will be given on DAY 2 (to allow drug interaction assessment).

# Appendix 2 Pharmacokinetic Sampling for Phase I, Metastatic Breast and Gastric Cancer Patients

| | Trastuzumab emtansine<br>(T-DM1), total<br>trastuzumab and DM1 <sup>a</sup><br>PK samples | Capecitabine and 5-FU<br>PK samples |
|---|---|---|
| Cycle 1 Day 1 | | |
| Pre-capecitabine dose | | Х |
| 30 min post capecitabine dosing | | X |
| 60 min post capecitabine dosing | | X |
| 1.5 hours post capecitabine dosing | | X |
| 2 hours post capecitabine dosing | | х |
| 2.5 hours post capecitabine dosing | | х |
| 4 hours post capecitabine dosing | | х |
| 6 hours post capecitabine dosing | | х |
| Cycle 1 Day 2 | | |
| Pre-T-DM1 dose | Х | |
| 15-30 min after end of T-DM1infusion | х | |
| Pre-capecitabine dose | | X |
| 30 min post capecitabine dosing | | X |
| 2 hours post capecitabine dosing | | X |
| 6 hours post capecitabine dosing | | х |
| Cycle 1 Day 3 | | |
| 24 hours (± 2 hours) after the end of infusion of T-DM1 | х | |
| Cycle 1 Day 8 | | |
| 7 days (± 1 day) after the end of infusion of T-DM1 <sup>a</sup> | х | |
| Cycle 2 Day 1 | | |
| Pre- capecitabine and T-DM1 dose <sup>a</sup> | х | |
| 15–30 min after end of trastuzumab emtansine infusion | х | |
| 30 min post capecitabine dosing | | X |
| 60 min post capecitabine dosing | | Х |

### Trastuzumab emtansine—F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 2, 03 September 2013

| 1.5 hours post capecitabine dosing | | х |
|------------------------------------------------------------------|---|---|
| 2 hours post capecitabine dosing | | х |
| 2.5 hours post capecitabine dosing | | х |
| 4 hours post capecitabine dosing | | х |
| 6 hours post capecitabine dosing | | х |
| Cycle 2 Day 2 | | |
| 24 hours (± 2 hours) after the end of infusion of T-DM1 | х | |
| Cycle 2 Day 7 | | |
| 7 days (± 1 day) after the end of infusion of T-DM1 <sup>a</sup> | х | |
| Cycle 3 | | |
| Pre T-DM1 dose | Х | |

PK = pharmacokinetic; 5-FU = 5-fluoruracil

Data from historic studies have determined that results are the lower limit of quantitation.

<sup>&</sup>lt;sup>a</sup> = Plasma DM1 samples will not be collected at Day 7 post-infusion of T-DM1 neither at pre-dose of Cycle 2 and Cycle 3.

Selected sections from the Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1,<sup>1</sup> are presented below, with slight modifications and the addition of explanatory text as needed for clarity.<sup>2</sup>

### Measurability of Tumor at Baseline

#### **Definitions**

At baseline, tumor lesions/lymph nodes will be categorized as measurable or non-measurable as described below.

#### a. Measurable Tumor Lesions

**Tumor Lesions.** Tumor lesions must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size as follows:

- 10 mm by CT or magnetic resonance imaging (MRI) scan (CT/MRI scan slice thickness/interval no greater than 5 mm)
- 10mm caliper measurement by clinical examination (lesions that cannot be accurately measured with calipers should be recorded as nonmeasurable)
- 20 mm by chest X-ray

Malignant Lymph Nodes. To be considered pathologically enlarged and measurable, a lymph node must be ≥ 15 mm in the short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and follow-up, only the short axis will be measured and followed. See also notes below on "Baseline Documentation of Target and Non-Target Lesions" for information on lymph node measurement.

<sup>&</sup>lt;sup>1</sup> Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (Version 1.1). Eur J Cancer 2009;45:228–47.

<sup>&</sup>lt;sup>2</sup> For consistency within this document, the section numbers and cross-references to other sections within the article have been deleted and minor formatting changes have been made.

#### b. Non-Measurable Tumor Lesions

Non-measurable tumor lesions encompass small lesions (longest diameter > 10 mm or pathological lymph nodes with short axis ≥ 10 but < 15 mm) as well as truly non-measurable lesions. Lesions considered truly non-measurable include leptomeningeal disease, ascites, pleural or pericardial effusion, inflammatory breast disease, lymphangitic involvement of skin or lung, peritoneal spread, and abdominal mass/abdominal organomegaly identified by physical examination that is not measurable by reproducible imaging techniques.

### c. Special Considerations Regarding Lesion Measurability

Bone lesions, cystic lesions, and lesions previously treated with local therapy require particular comment, as outlined below.

#### Bone Lesions:

- Bone scan, PET scan, or plain films are not considered adequate imaging techniques for measuring bone lesions. However, these techniques can be used to confirm the presence or disappearance of bone lesions.
- Lytic bone lesions or mixed lytic-blastic lesions, with identifiable soft tissue components, that can be evaluated by cross-sectional imaging techniques such as CT or MRI can be considered as measurable lesions if the soft tissue component meets the definition of measurability described above.
- Blastic bone lesions are non-measurable.

#### Cystic Lesions:

- Lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor non-measurable) since they are, by definition, simple cysts.
- Cystic lesions thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of measurability described above. However, if non-cystic lesions are present in the same patient, these are preferred for selection as target lesions.

### Lesions with Prior Local Treatment:

 Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion. Study protocols should detail the conditions under which such lesions would be considered measurable.

### **Target Lesions: Specifications by Methods of Measurements**

#### a. Measurement of Lesions

All measurements should be recorded in metric notation, using calipers if clinically assessed. All baseline evaluations should be performed as close as possible to the treatment start and never more than 28 days before the beginning of the treatment.

#### b. Method of Assessment

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during the study. Imaging-based evaluation should always be the preferred option.

**Clinical Lesions.** Clinical lesions will only be considered measurable when they are superficial and ≥ 10 mm in diameter as assessed using calipers (e.g., skin nodules). For the case of skin lesions, documentation by color photography including a ruler to estimate the size of the lesion is suggested.

**Chest X-Ray.** Chest CT is preferred over chest X-ray, particularly when progression is an important endpoint, since CT is more sensitive than X-ray, particularly in identifying new lesions. However, lesions on chest X-ray may be considered measurable if they are clearly defined and surrounded by aerated lung.

**CT, MRI.** CT is the best currently available and reproducible method to measure lesions selected for response assessment. This guideline has defined measurability of lesions on CT scan based on the assumption that CT slice thickness is 5 mm or less. When CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness. MRI is also acceptable.

If prior to enrollment it is known that a patient is unable to undergo CT scans with IV contrast because of allergy or renal insufficiency, the decision as to whether a non-contrast CT or MRI (without IV contrast) will be used to evaluate the patient at baseline and during the study should be guided by the tumor type under investigation and the anatomic location of the disease. For patients who develop contraindications to contrast after baseline contrast CT is done, the decision as to whether non-contrast CT or MRI (enhanced or non-enhanced) will be performed should also be based on the tumor type and the anatomic location of the disease, and should be optimized to allow for comparison with the prior studies if possible. Each case should be discussed with the radiologist to determine if substitution of these other approaches is possible and, if not, the patient should be considered not evaluable from that point forward. Care must

be taken in measurement of target lesions on a different modality and interpretation of non-target disease or new lesions, since the same lesion may appear to have a different size using a new modality.

**Ultrasound.** Ultrasound is not useful in assessment of lesion size and should not be used as a method of measurement.

**Endoscopy, Laparoscopy, Tumor Markers, Cytology, Histology.** The utilization of these techniques for objective tumor evaluation cannot generally be advised.

### **Tumor Response Evaluation**

#### **Assessment of Overall Tumor Burden and Measurable Disease**

To assess objective response or future progression, it is necessary to estimate the overall tumor burden at baseline and use this as a comparator for subsequent measurements. Measurable disease is defined by the presence of at least one measurable lesion, as detailed above.

### **Baseline Documentation of Target and Non-Target Lesions**

When more than one measurable lesion is present at baseline, all lesions up to a maximum of five lesions total (and a maximum of two lesions per organ) representative of all involved organs should be identified as target lesions and will be recorded and measured at baseline. This means that, for instances in which patients have only one or two organ sites involved, a maximum of two lesions (one site) and four lesions (two sites), respectively, will be recorded. Other lesions (albeit measurable) in those organs will be recorded as non-measurable lesions (even if the size is > 10 mm by CT scan).

Target lesions should be selected on the basis of their size (lesions with the longest diameter) and be representative of all involved organs, but in addition should lend themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion does not lend itself to reproducible measurement, in which circumstance the next largest lesion that can be measured reproducibly should be selected.

Lymph nodes merit special mention since they are normal anatomical structures that may be visible by imaging even if not involved by tumor. As noted above, pathological nodes that are defined as measurable and may be identified as target lesions must meet the criterion of a short axis of  $\geq$  15 mm by CT scan. Only the short axis of these nodes will contribute to the baseline sum. The short axis of the node is the diameter normally used by radiologists

to judge if a node is involved by solid tumor. Nodal size is normally reported as two dimensions in the plane in which the image is obtained (for CT this is almost always the axial plane; for MRI the plane of acquisition may be axial, sagittal, or coronal). The smaller of these measures is the short axis. For example, an abdominal node that is reported as being 20 mm × 30 mm has a short axis of 20 mm and qualifies as a malignant, measurable node. In this example, 20 mm should be recorded as the node measurement. All other pathological nodes (those with short axis ≥ 10 mm but < 15 mm) should be considered non-target lesions. Nodes that have a short axis of < 10 mm are considered non-pathological and should not be recorded or followed.

A sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the baseline sum of diameters. If lymph nodes are to be included in the sum, then, as noted above, only the short axis is added into the sum. The baseline sum of diameters will be used as a reference to further characterize any objective tumor regression in the measurable dimension of the disease.

All other lesions (or sites of disease), including pathological lymph nodes, should be identified as non-target lesions and should also be recorded at baseline. Measurements are not required and these lesions should be followed as "present," "absent," or in rare cases "unequivocal progression."

In addition, it is possible to record multiple non-target lesions involving the same organ as a single item on the Case Report Form (CRF) (e.g., "multiple enlarged pelvic lymph nodes" or "multiple liver metastases").

### Response Criteria

### a. Evaluation of Target Lesions

This section provides the definitions of the criteria used to determine objective tumor response for target lesions.

- Complete response (CR): Disappearance of all target lesions
   Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.</li>
- Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters
- Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline

In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.

The appearance of one or more new lesions is also considered progression.

 Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study

### b. Special Notes on the Assessment of Target Lesions

**Lymph Nodes.** Lymph nodes identified as target lesions should always have the actual short axis measurement recorded (measured in the same anatomical plane as the baseline examination), even if the nodes regress to < 10 mm on study. This means that when lymph nodes are included as target lesions, the sum of lesions may not be zero even if CR criteria are met, since a normal lymph node is defined as having a short axis of < 10 mm.

Target Lesions That Become Too Small to Measure. During the study, all lesions (nodal and non-nodal) recorded at baseline should have their actual measurements recorded at each subsequent evaluation, even when very small (e.g., 2 mm). However, sometimes lesions or lymph nodes that are recorded as target lesions at baseline become so faint on CT scan that the radiologist may not feel comfortable assigning an exact measure and may report them as being too small to measure. When this occurs, it is important that a value be recorded on the CRF, as follows:

- If it is the opinion of the radiologist that the lesion has likely disappeared, the measurement should be recorded as 0 mm.
- If the lesion is believed to be present and is faintly seen but too small to measure, a default value of 5 mm should be assigned and below measurable limit (BML) should be ticked. (Note: It is less likely that this rule will be used for lymph nodes since they usually have a definable size when normal and are frequently surrounded by fat such as in the retroperitoneum; however, if a lymph node is believed to be present and is faintly seen but too small to measure, a default value of 5 mm should be assigned in this circumstance as well and BML should also be ticked).

To reiterate, however, if the radiologist is able to provide an actual measure, that should be recorded, even if it is below 5 mm, and in that case BML should not be ticked.

**Lesions That Split or Coalesce on Treatment.** When non-nodal lesions fragment, the longest diameters of the fragmented portions should be added

together to calculate the target lesion sum. Similarly, as lesions coalesce, a plane between them may be maintained that would aid in obtaining maximal diameter measurements of each individual lesion. If the lesions have truly coalesced such that they are no longer separable, the vector of the longest diameter in this instance should be the maximum longest diameter for the coalesced lesion.

### c. Evaluation of Non-Target Lesions

This section provides the definitions of the criteria used to determine the tumor response for the group of non-target lesions. While some non-target lesions may actually be measurable, they need not be measured and instead should be assessed only qualitatively at the time points specified in the protocol.

- Complete response (CR): Disappearance of all non-target lesions and (if applicable) normalization of tumor marker level
  - All lymph nodes must be non-pathological in size (< 10 mm short axis).
- Non-CR/Non-PD: Persistence of one or more non-target lesions and/or (if applicable) maintenance of tumor marker level above the normal limits
- Progressive disease (PD): Unequivocal progression of existing non-target lesions

The appearance of one or more new lesions is also considered progression.

#### d. Special Notes on Assessment of Progression of Non-Target Disease

When the Patient Also Has Measurable Disease. In this setting, to achieve unequivocal progression on the basis of the non-target disease, there must be an overall level of substantial worsening in non-target disease in a magnitude that, even in the presence of SD or PR in target disease, the overall tumor burden has increased sufficiently to merit discontinuation of therapy. A modest increase in the size of one or more non-target lesions is usually not sufficient to qualify for unequivocal progression status. The designation of overall progression solely on the basis of change in non-target disease in the face of SD or PR of target disease will therefore be extremely rare.

When the Patient Has Only Non-Measurable Disease. This circumstance arises in some Phase III trials when it is not a criterion of study entry to have measurable disease. The same general concepts apply here as noted above; however, in this instance there is no measurable disease assessment to factor into the interpretation of an increase in non-measurable disease burden. Because worsening in non-target disease cannot be easily quantified (by definition: if all lesions are truly non-measurable), a useful test that can be

applied when assessing patients for unequivocal progression is to consider if the increase in overall disease burden based on the change in non-measurable disease is comparable in magnitude to the increase that would be required to declare PD for measurable disease, that is, an increase in tumor burden representing an additional 73% increase in volume (which is equivalent to a 20% increase in diameter in a measurable lesion). Examples include an increase in a pleural effusion from "trace" to "large" or an increase in lymphangitic disease from localized to widespread, or may be described in protocols as "sufficient to require a change in therapy." If unequivocal progression is seen, the patient should be considered to have had overall PD at that point. While it would be ideal to have objective criteria to apply to non-measurable disease, the very nature of that disease makes it impossible to do so; therefore, the increase must be substantial.

#### e. New Lesions

The appearance of new malignant lesions denotes disease progression; therefore, some comments on detection of new lesions are important. There are no specific criteria for the identification of new radiographic lesions; however, the finding of a new lesion should be unequivocal, that is, not attributable to differences in scanning technique, change in imaging modality, or findings thought to represent something other than tumor (e.g., some "new" bone lesions may be simply healing or flare of pre-existing lesions). This is particularly important when the patient's baseline lesions show partial or CR. For example, necrosis of a liver lesion may be reported on a CT scan report as a "new" cystic lesion, which it is not.

A lesion identified during the study in an anatomical location that was not scanned at baseline is considered a new lesion and will indicate disease progression.

If a new lesion is equivocal, e.g., because of its small size, continued therapy and follow-up evaluation will clarify if it represents truly new disease. If repeat scans confirm there is definitely a new lesion, then progression should be declared using the date of the initial scan.

### **Evaluation of Response**

#### a. Time Point Response (Overall Response)

It is assumed that at each protocol-specified time point, a response assessment occurs. **Table 1** provides a summary of the overall response status calculation at each time point for patients who have measurable disease at baseline.

When patients have non-measurable (therefore non-target) disease only, **Table 2** is to be used.

Table 1 Time Point Response: Patients with Target Lesions (with or without Non-Target Lesions)

| Target Lesions | Non-Target Lesions | New Lesions | Overall Response |
|---|---|---|---|
| | CR | No | CR |
| CR | | | |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | NE |
| PD | Any | Yes or no | PD |
| Any | PD | Yes or no | PD |
| Any | Any | Yes | PD |

$$\label{eq:crossing} \begin{split} &\text{CR=complete response; NE=not evaluable; PD=progressive disease; PR=partial response; SD=stable disease.} \end{split}$$

Table 2 Time Point Response: Patients with Non-Target Lesions Only

| Non-Target Lesions | New Lesions | Overall Response |
|--------------------|-------------|------------------|
| | No | CR |
| CR | | |
| Non-CR/non-PD | No | Non-CR/non-PD a |
| Not all evaluated | No | NE |
| Unequivocal PD | Yes or no | PD |
| Any | Yes | PD |

CR=complete response; NE=not evaluable; PD=progressive disease.

a "Non-CR/non-PD" is preferred over "stable disease" for non-target disease since stable disease is increasingly used as an endpoint for assessment of efficacy in some trials; thus, assigning "stable disease" when no lesions can be measured is not advised.

### b. Missing Assessments and Not Evaluable Designation

When no imaging/measurement is done at all at a particular time point, the patient is not evaluable at that time point. If only a subset of lesion measurements are made at an assessment, usually the case is also considered not evaluable at that time point, unless a convincing argument can be made that the contribution of the individual missing lesion(s) would not change the assigned time point response. This would be most likely to happen in the case of PD. For example, if a patient had a baseline sum of 50 mm with three measured lesions and during the study only two lesions were assessed, but those gave a sum of 80 mm, the patient will have achieved PD status, regardless of the contribution of the missing lesion.

If one or more target lesions were not assessed either because the scan was not done or the scan could not be assessed because of poor image quality or obstructed view, the response for target lesions should be "unable to assess" since the patient is not evaluable. Similarly, if one or more non-target lesions are not assessed, the response for non-target lesions should be "unable to assess" except where there is clear progression. Overall response would be "unable to assess" if either the target response or the non-target response is "unable to assess" except where this is clear evidence of progression, as this equates with the case being not evaluable at that time point.

### c. Special Notes on Response Assessment

When nodal disease is included in the sum of target lesions and the nodes decrease to "normal" size (<10 mm), they may still have a measurement reported on scans. This measurement should be recorded even though the nodes are normal in order not to overstate progression should it be based on increase in size of the nodes. As noted earlier, this means that patients with CR may not have a total sum of "zero" on the CRF.

Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic deterioration." Every effort should be made to document objective progression even after discontinuation of treatment. Symptomatic deterioration is not a descriptor of an objective response; it is a reason for stopping study therapy. The objective response status of such patients is to be determined by evaluation of target and non-target disease as shown in **Table 1**, **Table 2**, **Table 3**.

Table 3 Best Overall Response When Confirmation Is Required

| Overall Response at First Time Point | Overall Response at | Post Overell Peanance |
|---|---|---|
| Time Point | Subsequent Time Point | Best Overall Response |
| | CR | CR |
| CR | | |
| CR | PR | SD, PD, or PR <sup>a</sup> |
| CR | SD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| CR | PD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| CR | NE | SD, provided minimum<br>duration for SD was met;<br>otherwise, NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| PR | NE | SD, provided minimum<br>duration for SD was met;<br>otherwise, NE |
| NE | NE | NE |

CR=complete response; NE=not evaluable; PD=progressive disease; PR=partial response; SD=stable disease.

<sup>&</sup>lt;sup>a</sup> If a CR is truly met at the first time point, any disease seen at a subsequent time point, even disease meeting PR criteria relative to baseline, qualifies as PD at that point (since disease must have reappeared after CR). Best response would depend on whether the minimum duration for SD was met. However, sometimes CR may be claimed when subsequent scans suggest small lesions were likely still present and in fact the patient had PR, not CR, at the first time point. Under these circumstances, the original CR should be changed to PR and the best response is PR.

For equivocal findings of progression (e.g., very small and uncertain new lesions; cystic changes or necrosis in existing lesions), treatment may continue until the next scheduled assessment. If at the next scheduled assessment, progression is confirmed, the date of progression should be the earlier date when progression was suspected.

In studies for which patients with advanced disease are eligible (i.e., primary disease still or partially present), the primary tumor should also be captured as a target or non-target lesion, as appropriate. This is to avoid an incorrect assessment of CR if the primary tumor is still present but not evaluated as a target or non-target lesion.

### Appendix 4 Instructions for Scans in the Event of Isotope Shortage

Two key suppliers of Tc-99m generators (Chalk River Reactor, Canada and High Flux Reactor, the Netherlands) are expected to close. Supplies from other reactor sources will be unable to meet the expected world-wide patient-care needs. As a result, significant shortages of Tc-99m are expected, and the instructions listed below should be followed:

- ECHO will be the preferred imaging modality over MUGA scans to evaluate cardiac function.
- Tc-99m bone scans should be obtained as part of the baseline tumor assessment in all patients and should be repeated to confirm a CR or if progression of existing bone lesions and/or the development of new bone lesions is clinically suspected.
  - If a bone scan cannot be performed at baseline or if the investigator suspects that a bone scan may not be able to be repeated during the course of the study because of the Tc-99m shortage, the investigator may choose F-18 NaF or FDG-PET scan as an alternative.
- If bone lesions are selected as index non-target lesions, they must be
  apparent on baseline CT scans or other radiographic modalities (e.g.,
  skeletal X-rays that can be repeated in subsequent tumor assessments).
  Additional scans may be obtained to follow clinically important bone
  lesions if not visualized on the chest, abdomen, or pelvic CT scan.

These measures are intended to ensure that the same method of assessment and the same imaging technique is used throughout the study for each patient. If there is a question regarding the choice of alternatives in the event that a standard bone scan cannot be obtained during screening and/or during the study, please contact the Medical Monitor.

## Appendix 5 New York Heart Association Classification of Functional Cardiac Capacity

| Class | |
|---|---|
| I | No limitation: Ordinary physical activity does not cause undue fatigue, dyspnea, or palpitation. |
| II | Slight limitation of physical activity: Such patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitations, dyspnea, or angina. |
| III | Marked limitation of physical activity: Although patients are comfortable at rest, less than ordinary physical activity will lead to symptoms. |
| IV | Inability to carry on physical activity without discomfort: Symptoms of congestive heart failure are present even at rest. With any physical activity, increased discomfort is experienced. |

From: Criteria Committee, New York Heart Association, Inc. Diseases of the heart and blood vessels. Nomenclature and criteria for diagnosis. 6th ed. Boston, Little, Brown and Co, 1964:114.

### Appendix 6 ECOG Performance Status

| | Scale |
|---|---|
| Grade | |
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, i.e., light housework, office work |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair |
| 5 | Dead |

http://www.ecog.org/general/perf\_stat.html

### Memo



| То: | To whom it concern | Protocol No: MO28230 |
|---------|-----------------------|----------------------|
| Copies: | PDR-CDC or equivalent | |
| From: | MO28230 SMT | |
| Date: | 22nd October 2013 | |

#### Protocol version 2: Correction of Inclusion Criterion 8d Liver function

This Note to File is in regards to the current protocol version 2 and protocol Sections 4.1.3.1 and 4.1.3.2: Inclusion Criterion 8d Liver function.

These sections currently define criteria 8 d) liver function as below:

Evidence of stable liver function during the month prior to enrollment with liver function tests' (LFTs) fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN.

Due to a typo error in protocol version 2, criteria 8 d) liver function should read as below:

Evidence of stable liver function during the month prior to enrollment with liver function tests' (LFTs) fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN

Investigators are asked to enroll patients only if patients show evidence of stable liver function during the month prior to enrollment with liver function tests' (LFTs) fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin), regardless of whether they have bones metastases.

All countries having submitted protocol version 2 to their regulatory authorities and/or IECs/IRBs are requested to submit this Note to file to their regulatory authorities (if local processes allow) and/or IECs/IRBs and investigators for information.





#### **PROTOCOL**

TITLE: PHASE I STUDY OF THE COMBINATION OF TRASTUZUMAB

EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY

ADVANCED/METASTATIC GASTRIC CANCER PATIENTS,

FOLLOWED BY A RANDOMIZED, OPEN-LABEL PHASE II STUDY OF TRASTUZUMAB EMTANSINE AND CAPECITABINE VERSUS

TRASTUZUMAB EMTANSINE ALONE IN HER2-POSITIVE

**METASTATIC BREAST CANCER** 

PROTOCOL NUMBER: MO28230 VERSION NUMBER: 3

**EUDRACT NUMBER:** 2012-001547-46


Capecitabine (RO091978)

MEDICAL MONITOR: MD

SPONSOR: F. Hoffmann-La Roche Ltd

DATE FINAL: Last date of signatures below

### FINAL PROTOCOL APPROVAL

Name
Date and signature

30 Jule 2014

Statistician

### CONFIDENTIAL STATEMENT

The information contained in this document, especially any unpublished data, is the property of F. Hoffmann-La Roche Ltd (or under its control) and therefore is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Ethics Committee or Institutional Review Board. It is understood that this information will not be disclosed to others without written authorization from Roche except to the extent necessary to obtain informed consent from persons to whom the drug may be administered.

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 3, 30 June 2014

### **TABLE OF CONTENTS**

| PR | OTOCOL ACC | CEPTANCE FORM | 10 |
|---|---|---|---|
| PR | OTOCOL SYN | NOPSIS | 11 |
| 1. | BACKGROU | IND | 28 |
| | 1.1 | Background on Disease | 28 |
| | 1.1.1 | HER2-Positive Breast Cancer | 28 |
| | 1.1.2<br>Gastric Ca | HER2-Positive Locally Advanced/Metastatic ncer | 29 |
| | 1.2 | Background on Study Drugs | 30 |
| | 1.2.1 | Trastuzumab Emtansine | 30 |
| | 1.2.1.1 | Study TDM3569g | 31 |
| | 1.2.1.2 | Study TDM4258g | 32 |
| | 1.2.1.3 | Study TDM4374g | 32 |
| | 1.2.1.4 | Study TDM4450g | 33 |
| | 1.2.1.5 | Study TDM4688g | 34 |
| | 1.2.1.6 | Phase III Study TDM4370g | 35 |
| | 1.2.1.7 | Phase III study TDM4997g | 35 |
| | 1.2.1.8 | Pharmacokinetics | 36 |
| | 1.2.2 | Capecitabine | 38 |
| | 1.2.2.1<br>Trastuz | Study BO18255: Capecitabine and zumab in LA/mGC | 39 |
| | 1.2.3<br>Trastuzum | Preclinical Data of the Combination of ab Emtansine and a Fluoropyrimidine | 40 |
| | 1.3 | Study Rationale and Risk-Benefit Assessment | 41 |
| | 1.3.1 | For mBC | 41 |
| | 1.3.2 | For mGC | 42 |
| 2. | OBJECTIVES | | 43 |
| | 2.1 | Phase I: MTD-Finding of Trastuzumab Emtansine and Capecitabine in mBC | 43 |
| | 2.1.1 | Primary Objective | 43 |
| | 2.1.2 | Secondary Objectives | 43 |
| | 2.2 | Randomized Phase II: Exploration of Efficacy and Safety in mBC | 43 |
| | 2.2.1 | Primary Objective | |
| | 2.2.2 | Secondary Objectives | |
| | | nsine—F. Hoffmann-La Roche Ltd<br>/ersion 3, 30 June 2014 | 2 |

3

| | 2.3 | Phase I: MTD Finding of Trastuzumab Emtansine and Capecitabine in LA/mGC | 44 |
|---|---|---|---|
| | 2.3.1 | Primary Objective | 44 |
| | 2.3.2 | Secondary Objectives | 44 |
| 3. | STUDY DES | IGN | 44 |
| | 3.1 | Description of Study | 44 |
| | 3.1.1 | Overview of Study Design | 44 |
| | 3.1.1.1<br>mBC | Overview of Phase I Design in Patients with 46 | |
| | | Overview of Phase II: Exploration of Efficacy fety in Patients with mBC | 48 |
| | 3.1.1.3<br>Patient | Overview of Phase I Design in LA/mGC s 49 | |
| | 3.1.1.4 | Number of Patients | 49 |
| | 3.1.1.5 | Number of Centers | 50 |
| | 3.1.2 | Steering Committee | 50 |
| | 3.1.3 | Independent Data Monitoring Committee | 50 |
| | 3.2 | End of Study | 50 |
| | 3.3 | Rationale for Study Design | 50 |
| | 3.3.1 | Rationale for Patient Group Selection | 50 |
| | 3.3.1.1 | Rationale for Phase I | 51 |
| | 3.3.1.2 | Rationale for Randomized Phase II | 52 |
| | 3.3.2<br>Selection | Rationale for Investigational Medicinal Dose 52 | |
| | 3.3.2.1 | In Patients with mBC | 52 |
| | 3.3.2.2 | In Patients with mGC | 52 |
| | 3.3.2.3 | Rationale for Duration of Treatment | 53 |
| | 3.3.3 | Pharmacokinetic Sampling Rationale | 53 |
| | 3.4 | Outcome Measures | 53 |
| | 3.4.1 | Phase I: mBC | 53 |
| | 3.4.1.1 | Primary Outcome Measure | 53 |
| | 3.4.1.2 | Secondary Outcome Measure | 53 |
| | 3.4.1.3 | Primary Safety Outcome Measure | 53 |
| | 3.4.1.4 | Secondary Safety Outcome Measures | 54 |
| | 3.4.1.5 | Pharmacokinetic Outcome Measures | 54 |
| | 3.4.2 | Randomized Phase II: Exploration of Efficacy | |
| Tras | • | in mBCsine—F. Hoffmann-La Roche Ltd | 54 |

Protocol MO28230, Version 3, 30 June 2014

| | 3.4.2.1 | Primary Efficacy Outcome Measure | . 54 |
|----|--------------------|-----------------------------------------|------|
| | 3.4.2.2 | Secondary Efficacy Outcome Measures | . 55 |
| | 3.4.2.3 | Primary Safety Outcome Measure | . 55 |
| | 3.4.2.4 | Secondary Safety Outcome Measures | . 55 |
| | 3.4.2.5 | Pharmacokinetic Outcome Measures | . 55 |
| | 3.4.3 | Phase I: LA/mGC | . 55 |
| | 3.4.3.1 | Primary Outcome Measure | . 55 |
| | 3.4.3.2 | Secondary Efficacy Outcome Measure | . 56 |
| | 3.4.3.3 | Secondary Safety Outcome Measures | . 56 |
| | 3.4.3.4 | Pharmacokinetic Outcome Measures | . 56 |
| 4. | MATERIALS | AND METHODS | . 57 |
| | 4.1 | Patients | . 57 |
| | 4.1.1 | Patients with mBC | . 57 |
| | 4.1.2 | LA/mGC Patients | . 57 |
| | 4.1.3 | Inclusion Criteria | . 57 |
| | 4.1.3.1 | For Patients with mBC | . 57 |
| | 4.1.3.2 | For Patients with LA/mGC | . 58 |
| | 4.1.4 | Exclusion Criteria | . 60 |
| | 4.1.4.1 | For Patients with mBC | . 60 |
| | 4.1.4.2 | For Patients with LA/mGC | . 62 |
| | 4.1.5 | Patient Replacement Policy | . 63 |
| | 4.2 | Method of Treatment Assignment | . 63 |
| | 4.3 | Study Treatment | . 63 |
| | 4.3.1 | Formulation, Packaging, and Handling | . 63 |
| | 4.3.1.1 | Trastuzumab Emtansine | . 63 |
| | 4.3.1.2 | Capecitabine | . 64 |
| | 4.3.2 | Dosage and Administration | . 65 |
| | 4.3.2.1 | For Patients with mBC | . 65 |
| | 4.3.2.2 | For Patients with LA/mGC | . 66 |
| | 4.3.3<br>Accountab | Investigational Medicinal Product ility | . 66 |
| | 4.3.4 | Post-trial Access to Extension Study | . 66 |
| | 4.4 | Concomitant And Excluded Therapies | . 67 |
| | 4.4.1 | Permitted Therapy | . 67 |
| | 4.4.2 | Prohibited Therapy | . 67 |

| | 4.5 | Study Assessments | 68 |
|---|---|---|---|
| | 4.5.1 | Description of Study Assessments | 68 |
| | 4.5.1.1 | Medical History and Demographic Data | 68 |
| | 4.5.1.2 | Vital Signs | 68 |
| | 4.5.1.3 | Physical Examinations | 69 |
| | 4.5.1.4 | Tumor and Response Evaluations | 69 |
| | 4.5.1.5 | Laboratory Assessments | 70 |
| | 4.5.1.6 | Electrocardiograms | 70 |
| | 4.5.1.7 | ECOG Performance Status | 70 |
| | 4.5.1.8 | ECHO/MUGA | 71 |
| | 4.5.2 | Timing of Study Assessments | 71 |
| | 4.5.2.1 | Screening and Pretreatment Assessments | 71 |
| | 4.5.2.2 | Assessments during Treatment | 72 |
| | 4.5.2.3<br>Termina | Assessments at Study Completion/Early ation Visit | 72 |
| | | Follow-up Assessments | |
| | 4.5.2.5 | Assessments at Unplanned Visits | 73 |
| | 4.6 | Patient and STUDY Discontinuation | |
| | 4.6.1 | Patient Discontinuation | 73 |
| | 4.6.2 | Study Discontinuation | 73 |
| 5. | ASSESSME | NT OF SAFETY | 74 |
| | 5.1 | Safety Plan | 74 |
| | 5.1.1<br>Emtansine | Risks Associated with Trastuzumab 74 | |
| | 5.1.1.1 | Cardiotoxicity | 74 |
| | 5.1.1.2 | Hematologic Toxicity (Thrombocytopenia) | 74 |
| | 5.1.1.3 | Hepatotoxicity | 75 |
| | 5.1.1.4 | Pulmonary Toxicity | 76 |
| | 5.1.1.5 | Infusion-related Reactions/Hypersensitivity | 76 |
| | 5.1.1.6 | Neurotoxicity | 76 |
| | 5.1.1.7 | Extravasation | 77 |
| | 5.1.1.8 | Trastuzumab Emtansine Dose Modification | 77 |
| | 5.1.2 | Risks Associated with Capecitabine | 77 |
| | 5.1.3<br>Emtansine | Risks Associated with Trastuzumab and Capecitabine Combination | 78 |
| | 5.1.4 | Definition of Dose-limiting Toxicity | 78 |
| | | nsine—F. Hoffmann-La Roche Ltd<br>/ersion 3, 30 June 2014 | 5 |

| 5.1.5 | Management of Specific Adverse Events | 79 |
|---|---|---|
| 5.1 | .5.1 Trastuzumab Emtansine Dose Modification | <b>7</b> 9 |
| | 5.1.5.1.1 Trastuzumab Emtansine Dose Modification for Thrombocytopenia | 80 |
| | 5.1.5.1.2 Trastuzumab Emtansine Dose Modification for Hepatotoxicity | 81 |
| | 5.1.5.1.3 Trastuzumab Emtansine Dose Modification for Neurotoxicity | 82 |
| | 5.1.5.1.4 Trastuzumab Emtansine Dose Modification for Cardiotoxicity | 82 |
| | 5.1.5.1.5 Trastuzumab Emtansine Dose Modification/Management for Infusion-related Reactions, Hypersensitivity Reactions | 84 |
| | 5.1.5.1.6 Trastuzumab Emtansine Dose Modification for Pulmonary Toxicity | 85 |
| | 5.1.5.1.7 Trastuzumab Emtansine Dose Modification for Extravasation | 85 |
| 5.1 | .5.2 Capecitabine Dosage Modification | 85 |
| 5.2 | Safety Parameters and Definitions | 86 |
| 5.2.1 | Adverse Events | 86 |
| 5.2.2<br>Repor | Serious Adverse Events (Immediately table to the Sponsor) | 87 |
| 5.2.3<br>Interes | Protocol-defined Events of Special st/Non-Serious Expedited Adverse Events | 87 |
| 5.2.4 | Pregnancy and Contraception | 88 |
| 5.3 | Methods and Timing for Capturing and Assessing Safety Parameters | 90 |
| 5.3.1 | Adverse Event Reporting Period | 91 |
| 5.3.2 | Eliciting Adverse Event Information | 91 |
| 5.3.3 | Assessment of Severity of Adverse Events | 91 |
| 5.3.4 | Assessment of Causality of Adverse Events | 92 |
| 5.3.5 | Procedures for Recording Adverse Events | 93 |
| 5.3 | 3.5.1 Diagnosis <i>versus</i> Signs and Symptoms | 94 |
| | 3.5.2 Adverse Events Occurring Secondary to<br>ner Events | 94 |
| 5.3 | 3.5.3 Persistent or Recurrent Adverse Events | 94 |
| 5.3 | 3.5.4 Abnormal Laboratory Values | 95 |
| 5.3 | 3.5.5 Deaths | 95 |
| 5.3 | 3.5.6 Pre-Existing Medical Conditions | 95 |
| | Emtansine—F. Hoffmann-La Roche Ltd<br>230, Version 3, 30 June 2014 | 6 |

| | 5.3.5.7 | Lack of Efficacy or Clinical Worsening | 96 |
|---|---|---|---|
| | 5.3.5.8 | Hospitalization or Prolonged Hospitalization | 96 |
| | 5.4 | Immediate Reporting Requirements from Investigator to the Sponsor | 96 |
| | 5.4.1 | Emergency Medical Contacts | 97 |
| | 5.4.2<br>Events and<br>Interest | Reporting Requirements for Serious Adverse d Non-serious Adverse Events of Special 97 | |
| | 5.4.3 | Reporting Requirements for Pregnancies | 97 |
| | 5.4.3.1 | Pregnancies in Female Patients | 97 |
| | 5.4.3.2<br>Patient | <b>9</b> | |
| | 5.4.3.3 | Abortions | 98 |
| | 5.4.3.4 | Congenital Anomalies/Birth Defects | 98 |
| | 5.5 | Follow-up of Patients after Adverse Events | 99 |
| | 5.5.1 | Investigator Follow-up | 99 |
| | 5.5.2 | Sponsor Follow-up | 99 |
| | 5.6 | Post-study Adverse Events | 99 |
| | 5.7 | Expedited Reporting to Health Authorities, Investigators, Institutional Review Boards, and Ethics Committees | 99 |
| 6. | STATISTICAL CONSIDERATIONS AND ANALYSIS PLAN | | 100 |
| | 6.1 | Determination of Sample Size | 101 |
| | 6.2 | Summaries of Conduct of Study | 102 |
| | 6.3 | Summaries of Treatment Group Comparability | 102 |
| | 6.4 | Efficacy Analyses | 103 |
| | 6.4.1 | Primary Efficacy Endpoint | 103 |
| | 6.4.2 | Secondary Efficacy Endpoints | 105 |
| | 6.5 | Safety Analyses | 106 |
| | 6.6 | Pharmacodynamic Analyses | 108 |
| | 6.7 | Pharmacokinetic Analyses | 108 |
| | 6.8 | Exploratory Analyses | 109 |
| | 6.9 | Interim Analyses | 109 |
| 7. | DATA COLL | ECTION AND MANAGEMENT | 110 |
| | 7.1 | Data Quality Assurance | 110 |
| | 72 | Electronic Case Report Forms | 110 |

**Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 3, 30 June 2014

| | 7.3 | Source Data Documentation | 110 |
|---|---|---|---|
| | 7.4 | Use of Computerized Systems | 111 |
| | 7.5 | Retention of Records | 111 |
| 8. | ETHICAL | CONSIDERATIONS | 112 |
| | 8.1 | Compliance with Laws and Regulations | 112 |
| | 8.2 | Informed Consent | 112 |
| | 8.3 | Institutional Review Board or Ethics Committee | 113 |
| | 8.4 | Confidentiality | 113 |
| | 8.5 | Financial Disclosure | 114 |
| 9. | | OCUMENTATION, MONITORING, AND TRATION | 114 |
| | 9.1 | Study Documentation | 114 |
| | 9.2 | Site Inspections | 114 |
| | 9.3 | Administrative Structure | 114 |
| | 9.4 | Publication of Data and Protection of Trade Secrets | 114 |
| | 9.5 | Protocol Amendments | 115 |
| 10. | REFERE | NCES | 116 |
| | | LIST OF TABLES | |
| Tab | le 1 | Cycle 1 Mean (s.d.) Pharmacokinetic Parameters for Trastuzumab Emtansine Following Trastuzumab | |
| Table 2 | | Emtansine Administration Every 3 Weeks and Weekly in Study TDM3569g Dose Reduction for Trastuzumab Emtansine (Patients | 37 |
| | | with mBC) | 80 |
| lab | le 3 | Dose Reductions for Trastuzumab Emtansine (Patients with mGC) | 80 |
| Table 4 | | Trastuzumab Emtansine Dose Modification: Total Serum | |
| Table 5 | | Trastuzumab Emtansine Dose Modification: Serum ALT | |
| Tab | le 6 | or AST Adverse Event Severity Grading Scale | |
| | le 7 | Guidance for Causal Attribution of Adverse Event/Serious Adverse Event | |

### **LIST OF FIGURES**

**Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 3, 30 June 2014
| Figure 1<br>Figure 2 | Molecular Structure of Trastuzumab Emtansine | |
|---|---|---|
| Figure 3 | Anti-tumor Activity of Trastuzumab Emtansine in | |
| | Combination with Capecitabine in NCI-N87 | |
| Figure 4 | Overview of Study Design | |
| Figure 5 | Overview of Phase I Dose Finding Study Design | 47 |
| Figure 6 | Algorithm for Continuation and Discontinuation of | |
| | Trastuzumab Emtansine Based on Left Ventricular | 0.4 |
| | Ejection Fraction Assessments in Patients | 04 |
| | LIST OF APPENDICES | |
| | LIST OF APPENDICES | |
| Appendix 1 | Schedule of Assessments | 120 |
| Appendix 2<br>Metastat | Pharmacokinetic Sampling for Phase I, ic Breast and Gastric Cancer Patients | 129 |
| Appendix 3 | Response Evaluation Criteria in Solid | |
| • • | (RECIST): Modified Excerpt from Original | |
| · · | on | 131 |
| Appendix 4 | Instructions for Scans in the Event of Isotope | |
| Shortage | · | 143 |
| Appendix 5 | New York Heart Association Classification of | |
| Function | al Cardiac Capacity | 144 |
| Appendix 6 | ECOG Performance Status | 145 |

## PROTOCOL ACCEPTANCE FORM

TITLE: PHASE I STUDY OF THE COMBINATION OF TRASTUZUMAB
EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE
METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY

METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED OR METASTATIC GASTRIC CANCER PATIENTS, FOLLOWED BY A RANDOMIZED, OPEN-LABEL PHASE II STUDY OF TRASTUZUMAB EMTANSINE AND CAPECITABINE VERSUS

TRASTUZUMAB EMTANSINE ALONE IN HER2-POSITIVE

METASTATIC BREAST CANCER


**EUDRACT NUMBER:** 2012-001547-46


Capecitabine (RO091978)

**MEDICAL MONITOR:** 

**SPONSOR:** F. Hoffmann-La Roche Ltd

I agree to conduct the study in accordance with the current protocol.

| Principal Investigator's Name (print) | |
|---------------------------------------|------|
| Principal Investigator's Signature | Date |

Please return the signed original of this form {as instructed by XX [e.g., your local study monitor, the CRO]} [or] {to the contact provided below}. Please retain

a copy for your study files.

{Name} {Address}

#### PROTOCOL SYNOPSIS

TITLE: PHASE I STUDY OF THE COMBINATION OF TRASTUZUMAB EMTANSINE
(T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST
CANCER AND HER2-POSITIVE LOCALLY ADVANCED/METASTATIC GASTRIC
CANCER PATIENTS, FOLLOWED BY A RANDOMIZED, OPEN-LABEL PHASE II

STUDY OF TRASTUZUMAB EMTANSINE AND CAPECITABINE VERSUS TRASTUZUMAB EMTANSINE ALONE IN HER2-POSITIVE METASTATIC


**EUDRACT NUMBER:** 2012-001547-46

**BREAST CANCER** 


Capecitabine (RO091978)

PHASE: I/I

INDICATION: HER2-positive metastatic breast cancer or HER2-positive locally

advanced/metastatic gastric cancer

SPONSOR: F. Hoffmann-La Roche Ltd

#### **Objectives**

## Phase I: Maximum Tolerated Dose (MTD) Finding of Trastuzumab Emtansine (T-DM1) and Capecitabine in Metastatic Breast Cancer (mBC)

## Primary Objective

 To determine the MTD of the combination of trastuzumab emtansine and capecitabine in patients with human epidermal growth factor receptor 2 (HER2)-positive mBC

#### Secondary Objectives

To assess the:

- Pharmacokinetics (PK) of trastuzumab emtansine, capecitabine, and their metabolites
- Safety of the combination of trastuzumab emtansine and capecitabine
- Overall response rate (ORR)

## Randomized Phase II: Exploration of Efficacy and Safety in mBC

#### Primary Objective

 To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone in patients with HER2-positive mBC, as measured by ORR by Response Evaluation Criteria for Solid Tumors (RECIST) v.1.1 per investigator local assessment

#### Secondary Objectives

- To assess the safety profile of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone
- To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone in mBC patients, as measured by:
  - Time to response (TTR)
  - Duration of response (DoR)
  - Time to progression (TTP)
  - Time to treatment failure (TTF)

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- Progression-free survival (PFS)
- · Clinical benefit rate (CBR)
- Overall survival (OS)

## Phase I: MTD Finding of Trastuzumab Emtansine and Capecitabine in Locally Advanced/Metastatic Gastric Cancer (LA/mGC)

#### **Primary Objective**

 To determine the MTD of the combination of trastuzumab emtansine and capecitabine in patients with LA/mGC

#### **Secondary Objectives**

To assess the:

- PK of trastuzumab emtansine, capecitabine, and their metabolites
- Safety of the combination of trastuzumab emtansine and capecitabine
- ORR

#### **Study Design**

#### **Description of Study**

This is an international, multicenter study.

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with HER2-positive mBC or LA/mGC using a Phase I design, followed by a randomized, open-label Phase II study to explore the efficacy and safety of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone in HER2-positive mBC. Results from the Phase I study in LA/mGC will be used as supporting information for future studies in the indication (see Figure 4 in the protocol).

## Phase I: MTD Finding, Cohort 1: mBC

Cohort 1 used a 3 plus 3 classical design to determine the MTD of capecitabine in combination with trastuzumab emtansine. Initially the study had a dose escalation design, but following the occurrence of two DLTs at Dose Level 1 (750 mg/m² capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine), the study design was adapted and the dose descalated to 700 mg/m² capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine. At this Dose Level there were no DLTs and following review of the safety data, the Independent Data Monitoring Committee (IDMC) recommended that the study should proceed to explore this Dose Level further in the Randomized Phase II part of the study.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

Phase II will be conducted in mBC patients only. This part of the study will explore the efficacy and safety of the combination treatment of trastuzumab emtansine (T-DM1) and capecitabine, at 700 mg/m² bid (the recommended MTD), compared with trastuzumab emtansine alone in patients with mBC.

Approximately 210 additional patients with HER2-positive mBC will be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to the Phase II part of the study; however, they will be followed up until end of study (EOS).

## Phase I: MTD Finding, Cohort 2: LA/mGC

Cohort 2 will have a 3 plus 3 classical design and enroll patients with HER2-positive LA/mGC. Trastuzumab emtansine will be administered weekly at a dose of 2.4 mg/kg and capecitabine will start at dose level -1 (700 mg/m², the MTD defined in Cohort 1), with deescalation if required as follows:

- If Dose Level -1 is well tolerated (DLT in ≤ 1/6 patients), this dose will be established as the MTD for LA/mGC
- If Dose Level -1 is not tolerated in Cohort 2 (DLT in > 1/6 patients), de-escalation will be to Dose Level -2.
- If Dose Level -2 is too toxic, the combination of capecitabine with trastuzumab emtansine 2.4 mg/kg every week may be considered unfeasible in LA/mGC, recruitment will be terminated and the LA/mGC part will be closed. However, this will have no impact on continuation of the Randomized Phase II mBC part.

## Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

#### **Duration of treatment and follow-up**

All patients will be treated until investigator-assessed disease progression, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor. If toxicity is considered by the investigator to be related to only one of the two agents, the non-implicated agent can be continued as single-agent therapy.

All patients will be followed up until withdrawal of consent, death, or for up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first.

#### **Number of Patients**

Phase I, Cohort 1: mBC

A minimum of 6 and up to 18 patients will be enrolled.

Randomized Phase II: Exploration of Efficacy and Safety in mBC

Exploration of efficacy and safety in mBC will be based on approximately 210 randomized patients in total.

Phase I, Cohort 2: LA/mGC

A total of 6 to 12 patients will be enrolled.

#### **Target Population**

Phase I, Cohort 1: mBC

Patients with HER2-positive mBC will be enrolled.

The patient's HER2 status will be considered positive if the local institution or reference lab reported immunohistochemistry (IHC) 3+ staining intensity (on a scale of 0 to 3) or *in situ* hybridization (ISH) positive.

The HER2 status will be retrospectively confirmed by IHC and/or ISH in a central laboratory using archival paraffin-embedded tumor tissue. Retrospective central confirmation will not affect the treatment decisions or primary endpoint of Phase I and will be used to validate efficacy analyses in Phase I.

Before entering the study, patients must have received at least one prior treatment regimen for early or metastatic disease, which included a chemotherapy agent and trastuzumab either separately or in combination.

Randomized Phase II: Exploration of Efficacy and Safety in mBC

Patients with HER2-positive mBC will be randomized to receive either the combination of trastuzumab emtansine with capecitabine or trastuzumab emtansine alone. Retrospective central confirmation will be used to categorize patients for subgroup analyses according to central HER2 testing.

Before entering the study, patients must have received at least one prior treatment regimen for early or metastatic disease, which included a chemotherapy agent and trastuzumab either separately or in combination.

#### Phase I, Cohort 2: LA/mGC

Patients with centrally confirmed HER2-positive LA/mGC will be enrolled.

Patients must not have received prior chemotherapy for advanced/metastatic disease.

#### Inclusion Criteria:

## For mBC Patients:

- 1. Male or female.
- 2. Age ≥ 18 years old.
- 3. Signed informed consent before any study-specific procedure.
- 4. Able and willing to comply with the protocol.
- 5. Negative serum pregnancy test for women of childbearing potential (including premenopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in the medical history confirming that the patient is not of childbearing potential.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- 6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 7 months after the last dose of study treatment (see Section 5.2.4 in the protocol).
- 7. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
- 8. Blood:
  - a) Platelet count > 100,000 cells/mm<sup>3</sup>
  - b) International normalized ratio (INR) < 1.5
  - c) Absolute neutrophil count (ANC) > 1,500 cells/mm<sup>3</sup>
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.

#### 9. Liver function:

- a) Total bilirubin  $\leq$  1.5 × upper limit of normal (ULN) or direct bilirubin  $\leq$  1.5 × ULN in patients with documented Gilbert's syndrome.
- b) Serum glutamic oxaloacetic transaminase (SGOT)/aspartate transaminase (AST) and serum glutamic pyruvic transaminase (SGPT)/alanine transaminase (ALT) ≤ 2.5 × ULN.
- c) Alkaline phosphatase ≤ 2.5 × ULN. In patients with bone metastases: alkaline phosphatase ≤ 5 × ULN.
- d) Evidence of stable liver function during the month prior to enrollment with liver function test (LFT) fluctuations not exceeding 2.5 × ULN (for AST, ALT) and 1.5 × ULN (for total bilirubin).

#### 10. Renal function:

a) Serum creatinine of < 177 μmol/L or calculated creatinine clearance (CL)</li>
 > 50 mL/min. If urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate ≤ 1 g of protein/24 hours.

## 11. Cardiac function:

- a) Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan.
- 12. Life expectancy ≥12 weeks
- 13. Histologically or cytologically confirmed breast cancer.
- 14. HER2-positive disease, defined as IHC 3+ or ISH positive.
- 15. Tumor block or 8 slides available for retrospective central confirmation of HER2-positivity (central confirmation not necessary for enrollment).
- 16. mBC with at least one measurable lesion according to RECIST v.1.1.
- 17. Disease progression on at least one prior regimen containing trastuzumab and chemotherapy either separately or in combination.
- 18. Patients must have recovered from previous treatments

#### For LA/mGC Patients:

- 1. Male or female
- 2. Age ≥ 18 years old.
- 3. Signed informed consent before any study-specific procedure.
- 4. Able and willing to comply with the protocol.
- 5. Negative serum pregnancy test for women of childbearing potential (including premenopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in the medical history confirming that the patient is not of childbearing potential.

343

- 6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 76 months after the last dose of study treatment (see Section 5.2.4 in the protocol).
- 7. ECOG performance status of 0, 1, or 2.
- 8. Blood:
  - a) Platelet count > 100,000 cells/mm<sup>3</sup>.
  - b) INR < 1.5.
  - c) ANC > 1,500 cells/mm<sup>3</sup>.
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 9. Liver function:
  - a) Total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤ 1.5 × ULN in patients with documented Gilbert's syndrome.
  - b) SGOT/AST and SGPT/ALT ≤ 2.5 × ULN.
  - c) Alkaline phosphatase ≤ 2.5 × ULN. In patients with bone metastases: alkaline phosphatase ≤ 5 × ULN.
  - d) Evidence of stable liver function during the month prior to enrollment with LFT fluctuations not exceeding 2.5 × ULN (for AST, ALT) and 1.5 × ULN (for total bilirubin).
- 10. Renal function:
  - a) Serum creatinine of < 177 μmol/L or calculated creatinine CL > 50 mL/min. If urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate ≤ 1 g of protein/24 hours.
- 11. Cardiac function:
  - a) LVEF ≥ 50% by ECHO or MUGA scan.
- 12. Life expectancy ≥12 weeks
- 13. Histologically or cytologically confirmed mGC or locally advanced GC.
- 14. HER2-positive tumor (primary tumor or metastatic lesion), defined as either IHC 3+ or IHC 2+ and ISH+, prospectively confirmed by a Sponsor-designated central laboratory prior to enrollment. ISH positivity is defined as a ratio of ≥ 2.0 for the number of HER2 gene copies to the number of signals for CEP17.
  - a) Archival tumor samples obtained from primary or metastatic sites are acceptable.
  - b) Invasive tumor for central confirmation of HER2 status is required.
  - c) A formalin-fixed paraffin-embedded (FFPE) tissue block with at least 5 mm of invasive tumor for central confirmation is preferred. If FFPE tissue blocks (or partial block) are unavailable due to country or site regulations, a minimum of 8 freshly cut unstained slides MUST be available for central review of HER2 status.
- Inoperable LA/mGC.

#### **Exclusion Criteria:**

#### For mBC Patients:

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or five half-lives, whichever is longer.
  - b) Hormonal therapy within 14 days.
  - c) Trastuzumab within 21 days.
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine.
- 3. Prior treatment with capecitabine.
- 4. History of severe or unexpected reactions to fluoropyrimidine or known hypersensitivity to fluorouracil.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogs, such as brivudine.
  - Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
  - Signs or symptoms suggesting that the patient has dihydropyrimidine dehydrogenase (DPD) deficiency.
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product.
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>.
  - b) Epirubicin > 900 mg/m<sup>2</sup>.
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control symptoms within 28 days before first study drug administration.
- Current peripheral neuropathy of Grade ≥ 3 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.4.0.
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above.
- 11. Current unstable ventricular arrhythmia requiring treatment.
- 12. History of symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] Classes II–IV).
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration.
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment.
- 15. Severe dyspnea at rest due to complications of advanced malignancy or currently requiring continuous oxygen therapy.
- 16. Clinically significant malabsorption syndrome or inability to take oral medication.
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease).
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment.
- 19. Current pregnancy or lactation.
- 20. Current known active infection with human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C virus (HBV/HCV).
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV deoxyribonucleic acid (DNA) viral load per local guidelines.
- 21. Lapatinib ≤ 14 days before first study drug administration.
- 22. Previous radiotherapy for the treatment of mBC is not allowed if:
  - a) The last fraction of radiotherapy has been administered within 14 days prior to first study drug administration (28 days for patients with radiotherapy to control symptoms of brain metastases, see exclusion criterion 8).
  - b) More than 25% of marrow-bearing bone has been irradiated.
  - c) Any acute toxicity has not resolved to Grade ≤ 1 before first study drug administration.

#### For LA/mGC Patients:

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half-lives, whichever is longer.

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

- b) Hormonal therapy within 14 days.
- c) Trastuzumab within 21 days.
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine.
- Prior treatment with capecitabine.
- 4. History of severe or unexpected reactions to fluoropyrimidine or known hypersensitivity to fluorouracil.
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogs, such as brivudine.
  - Rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
  - c) Signs or symptoms suggesting that the patient has DPD deficiency.
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product.
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>.
  - b) Epirubicin > 900 mg/m<sup>2</sup>.
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>.
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control symptoms within 28 days before first study drug administration.
- 9. Current peripheral neuropathy of Grade ≥ 3 according to NCI CTCAE, v4.0.
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above.
- 11. Current unstable ventricular arrhythmia requiring treatment.
- 12. History of symptomatic CHF (NYHA Classes II-IV).
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration.
- History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment.
- 15. Severe dyspnea at rest due to complications of advanced malignancy or currently requiring continuous oxygen therapy.
- 16. Clinically significant malabsorption syndrome or inability to take oral medication.
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation.
- 20. Current known active infection with HIV, HBV, and/or HCV
  - For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Previous chemotherapy for advanced/metastatic disease
  - a) Prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrollment into the study
- 22. Lapatinib ≤ 14 days before first study drug administration

### Length of Study

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to last 2 years in total (1 year for MTD Finding, 1 year for the Phase II Exploration of Efficacy and Safety in mBC).

#### **End of Study**

The study will end after the follow-up period has been completed as defined above. Last patient last visit (LPLV) is defined as the last data collection point, which can be either a clinic visit or a laboratory sample.

In case Dose Level -2 is too toxic in LA/mGC, the LA/mGC cohort may be terminated prematurely. Patients who, at that point, experience response according to RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent or with capecitabine, based on the risk-benefit balance and agreement with the SC.

Randomized Phase II Exploration of Efficacy and Safety in mBC: The primary analysis of best overall response (BOR) rate will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever occurs first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after randomization of the first patient. The EOS analysis (approximately 24 months after the last patient is randomized) will include an updated analysis of BOR, which will be done in a purely exploratory manner.

#### **Efficacy Outcome Measures**

Efficacy will be evaluated according to RECIST v.1.1.

- BOR rate
- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

## **Safety Outcome Measures**

- DLT assessment/determination of the MTD of capecitabine when combined with trastuzumab emtansine (Phase I only)
- Incidence, nature, and severity by NCI CTCAE v4.0 of adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation from either component of the study treatment, and AEs of special interest (AESIs)
- Fatal AEs and their causes
- Events to monitor
- · Laboratory parameters
- LVEF
- Treatment exposure
- Physical examinations
- Vital signs and ECOG performance status
- Premature withdrawal from study medication and/or study

## **Pharmacodynamic Outcome Measures**

Hospital visit parameters.

## Pharmacokinetic Outcome Measures

PK will be evaluated during Phase I for trastuzumab emtansine, capecitabine, and their metabolites (see Appendix 1, Schedule of Assessment in the protocol). In addition, PK samples may be taken *ad hoc*, in case of SAEs or unexpected toxicities, which may be suggestive of a potential drug-drug interaction.

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

#### **Investigational Medicinal Products**

#### For mBC Patients:

Trastuzumab emtansine will be administered q3w at a dose of 3.6 mg/kg intravenous (IV).

The total trastuzumab emtansine dose will be calculated based on the patient's weight on Day 1 of each cycle (or up to 3 days before) with no upper limit.

<u>Capecitabine</u> will be administered orally bid for 14 days followed by a 7-day rest period at the Dose Levels described in the 'Trial Design' section.

Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Rounding of the capecitabine dose, based on 150 mg and 500 mg tablet strength, will be allowed to the nearest target dose based on the patient's body surface area (BSA).

#### For LA/mGC Patients:

<u>Trastuzumab emtansine</u> will be administered on Day 1 of each 1-week cycle at a dose of 2.4 mg/kg IV.

The total trastuzumab emtansine dose will be calculated based on the patient's weight on Day 1 of each cycle (or up to 3 days before) with no upper limit.

<u>Capecitabine</u> will be administered orally bid for 14 days followed by a 7-day rest period at the Dose Levels -1 to -2 described in the 'Trial Design' section.

Capecitabine tablets should be swallowed with water within 30 minutes after a meal.

#### **Non-Investigational Medicinal Products**

Not applicable.

#### **Statistical Methods**

The study will include 2 phases and 2 cohorts:

- Phase I, Cohort 1: mBC MTD-Finding Cohort
- Randomized Phase II: Exploration of Efficacy and Safety in mBC
- Phase I, Cohort 2: LA/mGC MTD-Finding Cohort

Corresponding analyses as described in the protocol will be performed when all data from both study phases are collected and cleaned.

Randomized Phase II: The primary analysis of BOR will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever occurs first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after randomization of the first patient. The EOS analysis (approximately 24 months after the last patient is randomized) will include an updated analysis of BOR, which will be done in a purely exploratory manner.

#### Analysis of primary and secondary endpoints:

#### Analysis Populations:

Phase I, Cohort 1: MTD-Finding: mBC Patients

The main analysis population for DLT assessment is the DLT-evaluable population, which is defined as all enrolled and treated patients who have not experienced any major protocol violations (including violations of the inclusion and exclusion criteria) and have completed Cycle 1.

The safety population (SP) will include all patients who received at least one dose of study medication (trastuzumab emtansine and/or capecitabine) during Phase I.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

The main analysis population for the efficacy analysis will be the intent-to-treat (ITT) population, which will include all patients randomized in the Phase II part of the study. The per-protocol (PP) population will include all ITT patients who have at least one post-baseline tumor assessment during the Phase II part of the study and no major protocol violations, which will be defined in the statistical analysis plan (SAP).

The SP will include all patients who received at least one dose of study medication during the Randomized Phase II part of the study.

#### Phase I, Cohort 2: MTD-Finding, LA/mGC Patients

The main analysis population for DLT assessment is the DLT-evaluable population, which is defined as all enrolled and treated patients who have not experienced any major protocol

#### Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

violation (including violation of the inclusion and exclusion criteria) and have completed Cycle 1.

The SP will include all patients who received at least one dose of study medication during Phase I.

#### Efficacy Endpoints:

#### Phase I, Cohort 1: MTD-Finding, mBC

The primary objectives are defining the MTD and establishing the safety profile of the combination regimen.

ORR, as a main efficacy endpoint, will be assessed via BOR rate. The BOR is defined as the best response recorded from the date of enrollment until disease progression, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### Randomized Phase II: Exploration of Efficacy in mBC

The primary efficacy endpoint for the Phase II part of the study is the ORR, assessed via the BOR rate. BOR is defined as the best response recorded between randomization into the Phase II part of the study and disease progression, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. To be assigned a status of partial response (PR) or complete response (CR), i.e., to be a responder, changes in tumor measurements must be confirmed by repeated assessments performed no less than 28 days after the response criteria are first met, i.e., patients need to have two consecutive assessments of PR or CR.

The primary hypothesis of interest when comparing ORR – as assessed via BOR - between the two treatment groups, combination of trastuzumab emtansine and capecitabine *versus* trastuzumab emtansine alone:

- H0: π trastuzumab emtansine = π trastuzumab emtansine + capecitabine where π trastuzumab emtansine is BOR in trastuzumab emtansine alone and π trastuzumab emtansine + capecitabine is BOR in trastuzumab emtansine + capecitabine
- H1: π trastuzumab emtansine ≠ π trastuzumab emtansine + capecitabine

The number and proportions of responders and non-responders (based on BOR) together with the two-sided 90% Clopper-Pearson confidence intervals (Cls) will be presented for each treatment group. The difference in BOR between treatment groups will be displayed with associated 90% Cls using the Hauck-Anderson approach and p-value for the Fisher's exact test.

The secondary endpoints for the Phase II part of the study will be:

- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

Estimates for the survivor function of both treatment groups for TTR, DoR, TTP, TTF, PFS and OS will be obtained by using the Kaplan-Meier method. Hazard ratios and associated 90% CIs will be estimated from non-stratified and stratified (based on the stratification factor) Cox regression models.

CBR will include patients whose best (confirmed) response was PR or CR, or stable disease (SD) that lasted at least 6 months. CBR will be summarized in a similar way to the primary efficacy endpoint, ORR, as assessed by BOR.

Phase I, Cohort 2: MTD-Finding: LA/mGC

## Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

The primary objectives are defining the MTD and establishing the safety profile of the combination regimen.

Efficacy endpoints will be analyzed in a similar way to that described for Phase I, Cohort 1 in mBC.

#### Safety Endpoints:

#### Phase I, Cohort 1: MTD-Finding: mBC

The number and proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

Safety parameters for this study part will also be summarized by treatment dose. The summaries of AEs, SAEs, AEs that cause discontinuation from the study treatment, AESIs (as described in Section 5), and events to monitor will be analyzed in a similar way to AEs in Phase II. The summaries will include all patients who received at least one dose of study medication.

The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry will be presented in shift tables of NCI CTCAE grade at baseline *versus* worst grade during treatment for Phase I, Cohort 1.

LVEF over time will be summarized as mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications, and physical examinations, will be analyzed in a similar way. Exposure to study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in each category will be presented by bar charts at different time points.

#### Randomized Phase II: Exploration of Safety in mBC

Safety endpoints will be summarized by treatment group.

Safety endpoints during the Randomized Phase II part of the study will be assessed via: total AEs, Grade ≥ 3 AEs, SAEs, premature withdrawal from study medication, AESIs, events to monitor, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

The incidence of AEs and SAEs will be summarized according to the primary SOC and within each SOC, by MedDRA preferred term. Time to onset of the first episode of AESI will also be summarized via Kaplan-Meier method. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology, and biochemistry will be presented in shift tables of NCI CTCAE grade at baseline *versus* worst grade during treatment in the Randomized Phase II part of the study.

LVEF over time will be summarized as mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications, and physical examinations, will be analyzed in a similar way. Exposure to study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in each category will be presented by bar charts at different time points.

#### Phase I, Cohort 2: MTD-Finding: mGC

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

Safety parameters will be summarized in a similar way to that described for Phase I, Cohort 1 in mBC.

#### Pharmacokinetic Analysis

The following PK parameters of trastuzumab emtansine and capecitabine (not limited to these listed) will be determined only in the Phase I part of the study in all patients who receive study treatment using either non-compartmental and/or population methods, if data allow:

- Serum concentrations of trastuzumab emtansine (conjugate) and total trastuzumab
- Plasma concentrations of DM1, capecitabine, and its active metabolite 5-fluorouracil (5-FU)
- Total exposure (area under the serum concentration-time curve [AUC])
- Maximum concentration (C<sub>max</sub>)
- CL
- Volume of distribution (V<sub>d</sub>)
- Terminal half-life (T<sub>1/2</sub>)

All PK parameters will be listed and tabulated by treatment dose and by Cohort. Descriptive summary statistics including arithmetic mean, geometric mean (e.g., AUC and  $C_{\text{max}}$ ), median, range, standard deviation (s.d.), and coefficient of variation will be presented for each Cohort. Nonlinear mixed effects modeling will also be used; details will be presented in the SAP.

#### **Exploratory Analyses**

For all patients with mBC (Phase I, cohort 1; Phase II Exploration of Efficacy and Safety in mBC), a retrospective central confirmation of the HER2 status will be done. Further exploratory analyses will be done according to centrally confirmed HER2 status for selected endpoints, e.g. BOR and safety (AEs, SAEs, Grade ≥ 3 AEs, and AESIs).

Subgroup analysis for BOR, safety (AEs, SAEs, AEs with Grade ≥ 3, and AESIs) in the Randomized Phase II part of the study will be presented for both treatment groups with respect to: elderly *versus* younger patients; patients with ECOG 0–1 *versus* ECOG 2; and patients with ≤1 *versus* >1 prior treatment line for metastatic disease. More details will be presented in the SAP.

#### **Pharmacoeconomic Endpoint**

The number of hospital visits, number of days admitted, and type of visits (emergency department *versus* inpatient care) will be collected and compared. The reason for admission (disease progression *versus* AE) will also be assessed.

### **Determination of Sample Size**

## Sample Size for Phase I: MTD-Finding: mBC

This part will be based on a classical 3 plus 3 Phase I design. A minimum of 6 and up to 18 patients will be enrolled in Cohort 1. There is no formal sample size estimation for this part.

#### Sample Size for Randomized Phase II: Exploration of Efficacy and Safety in mBC

The sample size for the primary endpoint BOR is based on a Fisher's exact test with an alpha level of 5% (one-sided), power of 80% and the clinical assumption of a BOR rate of 43% with trastuzumab emtansine alone and 62.5% with the combination of trastuzumab emtansine and capecitabine. Approximately 210 patients (105 patients in each treatment group), including a 15% withdrawal rate, will be randomized with a 1:1 ratio to either trastuzumab emtansine alone or the combination of trastuzumab emtansine and capecitabine.

### **Stratification Factors**

The following stratification factor will be implemented in the Randomized Phase II part of the study:

 Number of prior lines of treatment for metastatic disease (≤1 or >1; excluding singleagent hormones).

A treatment line is defined as any treatment regimen given to a patient from treatment initiation until confirmed disease progression.

### Sample Size for Phase I, Cohort 2: MTD-Finding: LA/mGC

This part will be based on a classical 3 plus 3 Phase I design. Between 3 and 12 patients might be enrolled in Cohort 2. There is no formal sample size estimation for this part.

## Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

#### Interim analysis

There is no formal interim analysis of efficacy.

An independent data monitoring committee (IDMC) will recommend whether the Randomized Phase II part of the study can commence.

The IDMC will also monitor safety outcomes after 25, 75, and 150 patients have received at least 3 cycles of treatment (Cycle 3 Day 21) in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II part of the study or as requested.

Efficacy data will be provided only if required by the IDMC to estimate the risk-benefit balance for the patients. Further details on the function and logistics of the IDMC will be provided in the IDMC Charter.

## **LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS**

| Abbreviation | Definition |
|------------------|------------------------------------------------|
| ADL | activities of daily living |
| ADC | antibody-drug conjugate |
| AE | adverse event |
| AESI | adverse event of special interest |
| ALT | alanine transaminase |
| ANC | absolute neutrophil count |
| aPTT | activated partial thromboplastin time |
| ARDS | acute respiratory distress syndrome |
| AST | aspartate transaminase |
| AUC | area under the serum concentration-time curve |
| BC | breast cancer |
| bid | twice daily |
| BML | below measurable limit |
| BOR | best overall response |
| BSA | body surface area |
| BUN | blood urea nitrogen |
| CBR | clinical benefit rate |
| CHF | congestive heart failure |
| CI | confidence interval |
| CL | clearance |
| C <sub>max</sub> | maximum concentration |
| CR | complete response |
| CRO | contract research organization |
| CSR | clinical study report |
| СТ | computed tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DLT | dose-limiting toxicity |
| DM1 | derivative of maytansine |
| DoR | duration of response |
| DPD | dihydropyrimidine dehydrogenase |
| 5-DFUR | 5'-deoxy-5-fluorouridine |
| 5-FU | 5-fluorouracil |
| EC | Ethics Committee |
| ECG | electrocardiogram |
| ECHO | echocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

| EEA | European economic area |
|----------|-------------------------------------------------------------|
| EOS | end of study |
| EU | European Union |
| FDA | Food and Drug Administration |
| FFPE | formalin-fixed paraffin-embedded |
| FISH | fluorescence in situ hybridization |
| GC | gastric cancer |
| GCP | Good Clinical Practice |
| GEJ | gastroesophageal junction |
| HBV | hepatitis B virus |
| HCV | hepatitis C virus |
| HER | human epidermal growth factor receptor |
| HER2 | human epidermal growth factor receptor 2 |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | human immunodeficiency virus |
| HR | hazard ratio |
| ICH | International Conference on Harmonisation |
| IDMC | independent data monitoring committee |
| IgG | immunoglobulin |
| IHC | immunohistochemistry |
| ILD | interstitial lung disease |
| IMP | investigational medicinal product |
| IND | Investigational New Drug (application) |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| ISH | in situ hybridization |
| ITT | intent-to-treat |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| IxRS | interactive voice/web recognition system |
| LA/mGC | locally advanced/metastatic gastric cancer |
| LC-MS/MS | liquid chromatography electrospray tandem mass spectrometry |
| LFT | liver function test |
| LPLV | last patient last visit |
| LVEF | left ventricular ejection fraction |
| mBC | metastatic breast cancer |
| mGC | metastatic gastric cancer |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | magnetic resonance imaging |

| MTD | maximum tolerated dose |
|---|---|
| MUGA | multiple-gated acquisition |
| N | number of patients |
| NCI | National Cancer Institute |
| NE | not evaluable |
| NRH | nodular regenerative hyperplasia |
| NYHA | New York Heart Association |
| ORR | overall response rate |
| OS | overall survival |
| PD | progressive disease |
| PET | positron emission tomography |
| PFS | progression-free survival |
| PK | pharmacokinetic |
| PP | per-protocol |
| PR | partial response |
| PVC | polyvinyl chloride |
| QTcF | heart rate-corrected QT interval using the Fridericia formula |
| q3w | every 3 weeks |
| qw | weekly |
| RECIST | Response Evaluation Criteria for Solid Tumors |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SGOT | serum glutamic oxaloacetic transaminase |
| SC | Steering Committee |
| s.d. | standard deviation |
| SD | stable disease |
| SDV | source data verification |
| SGPT | serum glutamic pyruvic transaminase |
| SmPC | Summary of Product Characteristics |
| SOC | system-organ class |
| SP | safety population |
| SWFI | sterile water for injection |
| T <sub>1/2</sub> | terminal half-life |
| TTF | time to treatment failure |
| TTP | time to progression |
| TTR | time to response |
| ULN | upper limit of normal |
| V <sub>d</sub> | volume of distribution |
| V <sub>ss</sub> | volume of distribution at steady state |
| WBC | white blood cells |
| WHO | World Health Organization |
| astuzumah Emtansine—F I | Hoffmann-La Roche I td |

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

5-FU 5-fluorouracil

## 1. BACKGROUND

### 1.1 BACKGROUND ON DISEASE

## 1.1.1 HER2-Positive Breast Cancer

Breast cancer (BC) is the most common cancer in women worldwide, both in the developed and the developing world<sup>1</sup>, with an estimated 1.67 million new cases diagnosed in 2012. It is also the leading cause of cancer death in females in less developed regions, accounting for 324,000 deaths (14.3% of all cancer deaths) in 2012, and the second most common cause of cancer death in women in more developed regions (198,000 deaths, 15.4%) after lung cancer.<sup>1</sup> Metastatic breast cancer (mBC) is incurable, with the primary goal of treatment to extend life and palliate symptoms while preserving quality of life.

Human epidermal growth factor receptor 2 (HER2) is an important prognostic factor in BC and is a key factor influence treatment strategies. The human epidermal growth factor receptor (HER) tyrosine kinase receptor family comprises four receptors: HER1, HER2, HER3, and HER4. These receptors are important mediators of cell growth, survival, and differentiation.<sup>2</sup> Activation of HER receptors leads to receptor dimerization and cell signaling through the PI3-kinase/AKT pathway for promotion of tumor cell survival and through the mitogen-activated protein kinase pathway for cellular proliferation.

Overexpression of HER2 is observed in approximately 15–20% of human BCs. Several lines of scientific and clinical evidence support a direct role for HER2 overexpression in the aggressive growth and poor clinical outcomes associated with these tumors.<sup>3</sup> The development of trastuzumab in the 1990s provided women with HER2-overexpressing tumors with a markedly better outcome than was possible with chemotherapy alone. Increases in overall response rate (ORR), response duration, and progression-free survival (PFS) were associated with a 5-month overall survival (OS) advantage when trastuzumab was given in the first-line metastatic setting, as demonstrated in the initial Phase III trial.<sup>4</sup>

For patients with HER2-positive mBC, the combination of anti-HER2 therapy and a taxane is a globally accepted first-line treatment, based on the OS advantage demonstrated in three large pivotal trials.<sup>4–6</sup>

However, disease progresses in almost all patients with HER2-positive mBC and these patients require additional therapies. Importantly, such tumors continue to express high levels of HER2,<sup>7</sup> and neither the process of internalization nor the level of surface expression is altered when HER2 is bound by trastuzumab.<sup>8</sup>

After progression, the standard strategy is further HER2-directed therapy, either continuing trastuzumab with a different chemotherapy agent (eg trastuzumab plus capecitabine), or changing to a different HER2-directed regimen (eg lapatinib plus capecitabine). In a randomized Phase III trial,

GBG26, in patients whose disease had progressed on previous trastuzumab-containing therapy, the combination of trastuzumab and capecitabine was associated with significantly improved time to progression (TTP) (hazard ratio [HR] 0.69, median 8.2 *versus* 5.6 months, respectively) and ORR (48% *versus* 27%) compared with capecitabine alone. In another Phase III trial involving patients with advanced HER2-positive BC previously treated with an anthracycline, a taxane, and trastuzumab, the addition of lapatinib to capecitabine resulted in an increased ORR (24% *versus* 14%) and TTP (median 6.2 months *versus* 4.3 months) compared with capecitabine alone.

# 1.1.2 HER2-Positive Locally Advanced/Metastatic Gastric Cancer

Gastric cancer (GC) remains one of the most common malignancies in the world with an estimated 952,000 new cases in 2012. GC also continues to be a deadly disease; it is the third leading cause of cancer-related death, accounting for 723,000 deaths (8.8% of all cancer deaths) worldwide in 2012. The only potentially curative treatment for GC is complete resection of localized disease. The overall 5-year survival for all cases, regardless of initial stage at diagnosis, is less than 25%. The approximately 40–60% will have disease who undergo curative surgery, approximately 40–60% will have disease recurrence. Patients with unresectable disease due to locally advanced growth or metastatic spread have the poorest prognosis, with an overall 5-year survival rate in the range of 3% to 15%. The survival rate in the range of 3% to 15%. The survival rate in the range of 3% to 15%.

Whereas HER2 overexpression is associated with a poor prognosis in BC, the prognostic significance of HER2 overexpression in GC is not fully defined. Studies of HER2 positivity rates in GC have shown a broad variation of HER2 positivity ranging from 6.8% to 34.0% for immunohistochemistry (IHC) and 7.1% to 42.6% for fluorescence *in situ* hybridization (FISH) techniques. <sup>15,16</sup> In a recent study, HER2 positivity was shown in 17% of resected esophageal adenocarcinomas and was significantly associated with lower tumor grade, less invasiveness, fewer malignant nodes, and the presence of adjacent Barrett's esophagus. <sup>17</sup>

In the ToGA trial (study BO18255), a global, Phase III study of trastuzumab plus chemotherapy as first-line treatment for advanced HER2-positive GC, <sup>18</sup> an overall HER2-positivity rate of 22.1% was observed (810/3667 evaluable samples), which is similar to BC. A higher HER2 positivity rate was seen in adenocarcinoma of the gastroesophageal junction (GEJ) than in the stomach (33.2% *versus* 20.9%), and intestinal type GCs showed a significantly higher HER2 positivity rate than diffuse or mixed-type tumors (intestinal: 32.2%, diffuse: 6.1%, mixed: 20.4%).<sup>19</sup>

In the ToGA trial, the addition of trastuzumab to chemotherapy (capecitabine or fluorouracil combined with cisplatin) for the treatment of patients with HER2-positive (defined as IHC 3+ or FISH positive), inoperable, locally advanced or recurrent and/or metastatic adenocarcinoma of the stomach or GEJ resulted in an increase in OS (median 13.8 months *versus* 11.1 months, HR 0.74, p = 0.0046), ORR (47% *versus* 35%), PFS (median 6.7 *versus* 5.5

months), and TTP (median 7.1 versus 5.6 months) compared with chemotherapy alone.18

#### 1.2 BACKGROUND ON STUDY DRUGS

#### 1.2.1 TRASTUZUMAB EMTANSINE

Trastuzumab emtansine (Figure 1) is a novel antibody-drug conjugate (ADC) that is specifically designed for the treatment of HER2-positive malignancies. Trastuzumab emtansine is composed of: trastuzumab, a humanized monoclonal antibody directed against the extracellular region of HER2; an average of 3.5 molecules of derivative of maytansine (DM1; maytansinoid), an anti-microtubule agent; and the thioether linker maleimidylmethyl cylcohexane-1-carboxylate, which is used to conjugate each molecule of DM1 to trastuzumab. DM1 is a highly potent drug synthesized from maytansinol that binds β tubulin to inhibit tubulin polymerization. It binds to tubulin competitively with vinca alkaloids, but is 20-100 times more potent than vincristine in its cytotoxic effect against tumor cell lines. Its parent molecule, maytansine, was studied in approximately 800 cancer patients in the 1970s and 1980s, with responses seen in patients with breast and lung cancers.<sup>20,21</sup> However, because of its narrow therapeutic index and the observed gastrointestinal toxicity of the free drug, it was not developed further as a therapeutic option. 22,23

Figure 1 Molecular Structure of Trastuzumab Emtansine



~150,000 Ratio: 3.5 3.5 1

DM1 = Derivative of maytansine, a microtubule destabilizing agent MW = Molecular weight

738

Similar to trastuzumab, trastuzumab emtansine recognizes an epitope in the extracellular domain of HER2 and binds to HER2 with a similar affinity.

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 3, 30 June 2014

MW:

30

238

Following antigen-specific binding of trastuzumab emtansine to HER2, the complex of receptor and ADC is internalized, whereupon DM1-containing catabolites are released into the cytosol following proteolytic cleavage of the antibody in lysosomes. <sup>24</sup> Binding of these DM1-containing species to  $\beta$ -tubulin inhibits tubulin polymerization, resulting in cell death. <sup>22</sup>

In addition to targeting delivery of DM1 to HER2-overexpressing tumor cells, trastuzumab emtansine retains the anti-tumor activities of trastuzumab, including suppression of HER2 signaling pathways that confer a proliferative and survival advantage to cells, and the flagging of cells for destruction through antibody-dependent cell cytotoxicity.<sup>20</sup>

Phase I single-arm studies were conducted to identify the most appropriate dosing regimen for further clinical development, and assess the safety of trastuzumab emtansine. Low levels of DM1 in systemic circulation supported the stability of the linker. The studies also provided an indication of clinical activity and led to randomized evaluation of single-agent trastuzumab emtansine versus other HER2-directed therapy in combination with chemotherapy. These trials demonstrated significantly superior PFS and OS with trastuzumab emtansine. Ce-28

Data from clinical trials of trastuzumab emtansine that are relevant to the design of the current trial are summarized below. Please refer to the trastuzumab emtansine Investigator's Brochure for further information on all of the completed and ongoing trastuzumab emtansine studies.

## 1.2.1.1 Study TDM3569g

Study TDM3569g was a Phase I, dose-escalation study that evaluated the safety and efficacy of trastuzumab emtansine as a single agent in 52 patients with HER2-positive mBC, whose disease progressed on a trastuzumab-containing chemotherapy regimen.<sup>29,30</sup> The study was completed on 11 June 2009, with a total of 52 patients treated; 24 patients received trastuzumab emtansine every 3 weeks (q3w); 28 patients received trastuzumab emtansine on a weekly (qw) schedule.

On the q3w dosing schedule, dose-limiting toxicities (DLTs) of Grade 4 thrombocytopenia were seen in 2 of 3 patients treated at 4.8 mg/kg. Therefore, 3.6 mg/kg was determined to be the maximum tolerated dose (MTD) of trastuzumab emtansine given q3w, and the cohort was expanded to 15 patients. On the basis of these data, the recommended dose schedule for the Phase II studies was 3.6 mg/kg q3w. On the qw schedule, 2.4 mg/kg was identified as the MTD.

Treatment with trastuzumab emtansine was well tolerated, and toxicity was generally mild, reversible, and non-cumulative. No drug-related cardiac toxicity was noted.

Trastuzumab emtansine administration demonstrated considerable activity in this Phase I study. The confirmed ORR in patients with measurable disease at the 3.6 mg/kg q3w schedule was 44% (4 of 9 patients), as assessed by

investigators. The median PFS among the 15 patients receiving 3.6 mg/kg q3w was 10.4 months.

## 1.2.1.2 Study TDM4258g

Study TDM4258g was a Phase II study that evaluated the safety and efficacy of trastuzumab emtansine administered at a dose of 3.6 mg/kg (intravenous; IV) q3w in patients with HER2-positive mBC whose disease had progressed on previous HER2-directed therapy and conventional chemotherapy.<sup>31</sup>

The primary objectives for this study were: 1) to assess the ORR (by independent radiologic review) associated with trastuzumab emtansine 3.6 mg/kg IV q3w; and 2) to characterize the safety and tolerability of trastuzumab emtansine at this dose.

The study was activated on 20 July 2007, and enrollment was completed (n = 112) on 31 July 2008. The final analysis of ORR was performed with a data cut-off date of 25 June 2009, 11 months after the last patient was enrolled. The reported ORR in all patients was 37.5% (95% confidence interval [CI]: 28.6%–46.6%) by investigator assessment and 25.9% (95% CI: 18.4%–34.4%) by independent review. The clinical benefit rate (CBR; defined as complete response [CR], partial response [PR], or stable disease [SD] for >6 months) was 46.3% by investigator assessment and 39.3% by independent review. The median PFS was 4.6 months as assessed by both the investigators and independent review. In the subset of patients whose archival primary tumors were retrospectively confirmed to be HER2-positive (74 of 95 patients with submitted tumor samples), the ORR was 33.8% by independent review and 47.3% based on investigator assessment.

The most common adverse events (AEs) (occurring in  $\geq$  20% of patients) were fatigue (65.2%), nausea (50.9%), headache (40.2%), epistaxis (35.7%), pyrexia (34.8%), constipation (30.4%), cough (27.7%), hypokalemia (26.8%), diarrhea (25.9%), vomiting (24.1%), arthralgia (22.3%), pain in extremity (22.3%), anemia (20.5%), and dyspnea (20.5%). Most of these AEs were Grade 1–2. The three most common Grade 3–4 AEs observed in this trial were hypokalemia (8.9%), thrombocytopenia (8.0%), and fatigue (4.5%). There was one reported Grade 5 event in a patient who died of respiratory failure attributed by the investigator to underlying disease. No Grade  $\geq$  3 left ventricular systolic dysfunction events (symptomatic congestive heart failure [CHF] and/or left ventricular ejection fraction [LVEF] of < 40%) were observed.

## 1.2.1.3 Study TDM4374g

Study TDM4374g was a Phase II, single-arm study of trastuzumab emtansine administered at 3.6 mg/kg by IV infusion q3w to patients with HER2-positive mBC. Patients must have received an anthracycline, trastuzumab, a taxane, lapatinib, and capecitabine given in the neoadjuvant, adjuvant, or metastatic setting or as treatment for locally advanced disease. Patients must have been treated with two HER2-directed therapies in the metastatic or locally advanced setting and have experienced progressive disease (PD) on their most recent treatment.

The primary objectives of this study were: 1) to assess the ORR as determined by an independent review using the modified Response Evaluation Criteria for Solid Tumors (RECIST) v. 1.0; and 2) to characterize the safety and tolerability of this trastuzumab emtansine regimen in the aforementioned patient population. The study was activated on 2 May 2008, and enrollment was complete on 2 April 2009. A total of 110 patients were enrolled and treated in the study.

An efficacy analysis (data cut-off date: 21 June 2010) with a median follow-up of 17.4 months demonstrated an ORR (CR or PR) of 34.5% (95% CI: 26.1%–43.9%; 38 of 110 patients) by independent review and 32.7% (95% CI: 24.1%–42.1%; 36 patients) by investigator assessment. The CBR was 48.2% by independent review and 46.4% by investigator assessment. The median duration of response (DoR) and median PFS by independent review was 7.2 months and 6.9 months, respectively. In the subset of patients whose archival primary tumors were retrospectively confirmed to be HER2-positive (80 of 95 patients with submitted tumor samples), the ORR was 41.3% by independent review and 40.0% based on investigator assessment.

The most common AEs (occurring in  $\geq$  20% of patients) were fatigue (61.8%), thrombocytopenia (38.2%), nausea (37.3%), increased aspartate transaminase (AST, 26.4%), constipation (23.6%), pyrexia (22.7%), epistaxis (22.7%), headache (21.8%), hypokalemia (20.9%), decreased appetite (20.9%), dry mouth (20.0%), and anemia (20.0%). Most of these AEs were Grade 1–2. Fifty-two patients (47.3%) experienced at least one Grade  $\geq$  3 AE, the most common being thrombocytopenia (9.1%) and fatigue (4.5%). Serious AEs (SAEs) were recorded in 28 patients (25.5%), the most common being cellulitis (3.6%), pyrexia (2.7%), and pneumonia (2.7%). There was one Grade 5 AE (hepatic dysfunction), which was recorded as possibly related to trastuzumab emtansine. The patient had pre-existing non-alcoholic fatty liver disease as well as multiple other comorbidities, including renal insufficiency.

### 1.2.1.4 Study TDM4450g

This was a randomized, multicenter, Phase II study of the efficacy and safety of trastuzumab emtansine *versus* trastuzumab plus docetaxel in patients with metastatic HER2-positive BC who had not received prior chemotherapy for metastatic disease. <sup>26</sup> This study completed enrollment in December 2009 (n = 137). The co-primary objectives were to assess the efficacy of trastuzumab emtansine compared with the combination of trastuzumab and docetaxel, as measured by PFS based on investigator tumor assessments, and to characterize the safety of trastuzumab emtansine compared with the combination of trastuzumab and docetaxel in this population. Secondary endpoints included ORR, OS, and DoR.

The data cut-off date was 15 November 2010. Seventy patients were randomized to the control arm and 67 patients to the trastuzumab emtansine arm. The median duration of follow-up was 13.5 months for the control arm and 13.8 months for the trastuzumab emtansine arm.

As of 15 November 2010, the median PFS was 14.2 months in the trastuzumab emtansine arm versus 9.2 months in the trastuzumab plus docetaxel arm. The HR for PFS was 0.594 (95% CI: 0.364-0.968; p = 0.0353). The ORR in the trastuzumab emtansine arm was 64.2% (95% CI: 51.8%-74.8%) compared with 58.0% (95% CI: 45.5%–69.2%) in the control arm (based on 69 evaluable patients). The CBR was 74.6% (95% CI: 63.2%-84.2%) in the trastuzumab emtansine arm versus 81.2% (95% CI: 70.7%-89.1%) in the trastuzumab plus docetaxel arm (based on 69 evaluable patients). Based on safety data analyzed at the data cut-off date, single-agent trastuzumab emtansine appears to have a favorable overall safety profile compared with trastuzumab and docetaxel as first-line therapy for mBC. The incidence of Grade ≥ 3 AEs in the control arm (89.4%; n = 66) was nearly twice that of trastuzumab emtansine (46.4%; n = 69). The rates of SAEs for both arms were similar (control arm 25.8% versus trastuzumab emtansine 18.8%). One patient in the trastuzumab emtansine group died as a result of an AE (sudden death). This patient was randomized to receive trastuzumab plus docetaxel but mistakenly received a single dose of 6 mg/kg trastuzumab emtansine instead of 6 mg/kg trastuzumab. One patient in the trastuzumab plus docetaxel group died due to cardiopulmonary failure. With respect to cardiotoxicity, based on local assessments of LVEF, trastuzumab emtansine was not associated with an increase in cardiotoxicity compared with trastuzumab plus docetaxel.

## 1.2.1.5 Study TDM4688g

The effect of trastuzumab emtansine (3.6 mg/kg q3w) on the QT interval in patients with HER2-positive recurrent locally advanced BC or mBC was evaluated in study TDM4688g. No meaningful effect of trastuzumab emtansine on the corrected QT interval was seen in these patients. At Cycle 1 Day 1, 15 minutes post-infusion, the baseline-adjusted mean heart rate-corrected QT interval using the Fridericia formula (QTcF) increased by 1.2 ms. By 60 minutes post-infusion, the baseline-adjusted mean QTcF interval decreased by 1.0 ms, and by Day 8 of Cycle 1 the baseline-adjusted mean QTcF interval decreased by 4.0 ms. By Cycle 3 Day 1, prior to trastuzumab emtansine infusion, the mean QTcF interval had reverted to baseline. Following the third infusion of trastuzumab emtansine, the baseline-adjusted mean QTcF interval at both the 15-minute and the 60-minute post-infusion time points was increased by 4.7 ms. No patient exhibited a mean change in QTcF interval from baseline exceeding 30 ms at any of the protocol-specified time points.

The relationship between trastuzumab emtansine pharmacokinetic (PK) and electrocardiogram (ECG) data was also assessed. While there appears to be a trend between trastuzumab emtansine drug concentration and its effect on QT interval, at the observed concentration ranges of trastuzumab emtansine, DM1, and total trastuzumab, there is reasonable assurance that the true increase in mean baseline-adjusted average QTcF does not exceed 5 ms. Moreover, because trastuzumab emtansine, total trastuzumab, and DM1 achieve steady state levels by Cycle 3, the likelihood of progressively longer QTcF with repeated trastuzumab emtansine dosing is low.

In this study, the ORR was 25.5% (95% CI: 15.2%–38.5%) as assessed by the investigator; no independent review was performed. The CBR was 39.2% (95% CI: 25.8%–53.1%), and the median PFS was 4.3 months (95% CI: 4.0–6.7).

## 1.2.1.6 Phase III Study TDM4370g

A randomized, open-label Phase III trial (TDM4370g; EMILIA) compared single-agent trastuzumab emtansine *versus* lapatinib and capecitabine in patients with HER2-positive locally advanced unresectable BC or mBC who had received a prior taxane and trastuzumab therapy and had documented PD.<sup>27</sup>

Patients were randomized in a 1:1 ratio to trastuzumab emtansine 3.6 mg/kg IV q3w or the combination of oral capecitabine 1,000 mg/m² twice daily (bid) on Days 1–14 q3w plus oral lapatinib 1,250 mg/day given as continuous dosing. Treatment was continued until PD (as assessed by the investigator), unmanageable toxicity, or study termination. PFS and OS were co-primary endpoints, with PFS based on modified RECIST³⁴ and assessed by independent review. Key secondary endpoints were ORR, DoR, and CBR, determined both by the investigator and by independent review.

The study demonstrated statistically significant and clinically meaningful improvements in both PFS and OS for trastuzumab emtansine compared with lapatinib plus capecitabine. Median PFS was 9.6 months in the trastuzumab emtansine arm *versus* 6.4 months in the control arm (HR = 0.65; 95% CI: 0.55–0.77; p < 0.001, log-rank test). Median OS was 30.9 months *versus* 25.1 months, respectively (HR = 0.68; 95% CI: 0.55–0.85; p < 0.001, log-rank test).

This benefit was supported by consistent improvements in all secondary efficacy endpoints, including investigator-assessed PFS, ORR, time to treatment failure (TTF), and the patient-reported outcome of time to symptom progression. The ORR in the trastuzumab emtansine arm was 43.6% (95% CI: 38.6%–48.6%) compared with 30.8% (95% CI: 26.3%–35.7%) in the control arm (based on 786 evaluable patients). Single-agent trastuzumab emtansine appears to have a favorable overall safety profile compared with lapatinib and capecitabine in mBC. The incidence of Grade  $\geq$  3 AEs in the control arm (56.9%; n = 488) was 278; that of trastuzumab emtansine (40.8%; n = 490) was 200. The rates of SAEs for both arms were similar (control arm 18% *versus* trastuzumab emtansine 15.5%).

Based on the results of this phase III trial, both the Food and Drug Administration (FDA) in the US and the European Commission in Europe approved trastuzumab emtansine for the treatment of HER2-positive mBC previously treated with trastuzumab and a taxane.

## 1.2.1.7 Phase III study TDM4997g

A second open-label randomized Phase III trial (TDM4997g; TH3RESA) compared single-agent trastuzumab emtansine *versus* the investigator's choice of therapy in patients with HER2-positive advanced BC who had previously received two or more HER2-directed regimens in the advanced

setting, including trastuzumab and lapatinib, and previous taxane therapy in any setting.<sup>28</sup> A total of 602 patients were randomized in a 2:1 ratio (404 to trastuzumab emtansine and 198 to physician's choice).

After median follow-up of approximately 7 months in both arms, 219 patients (54%) in the trastuzumab emtansine group and 129 (65%) in the physician's choice group had experienced PFS events. PFS was significantly improved with trastuzumab emtansine compared with physician's choice (HR 0.528, p<0.0001; median PFS 6.2 months with trastuzumab emtansine *versus* 3.3 months in the control arm. The HR for OS at the interim analysis was 0.552 (95% CI 0.369–0.826) but the stopping boundary was not crossed. Grade ≥3 AEs occurred less frequently with trastuzumab emtansine than with physician's choice (32% of patients vs 43%). Grade ≥3 neutropenia, diarrhea, and febrile neutropenia were less common with trastuzumab emtansine than physician's choice, whereas grade ≥3 thrombocytopenia (5% *vs* 2%) was more common with trastuzumab emtansine.

#### 1.2.1.8 Pharmacokinetics

The PK of trastuzumab emtansine and its analytes (total trastuzumab and DM1) were characterized in one Phase I study (TDM3569g) and three Phase II studies (TDM4258g, TDM4374g, and TDM4688g).

For study TDM3569g, the final PK parameter estimates based on non-compartmental PK analysis for q3w and qw regimens of trastuzumab emtansine administration are presented in Table 1.

Table 1 Cycle 1 Mean (s.d.) Pharmacokinetic Parameters for Trastuzumab Emtansine Following Trastuzumab Emtansine Administration q3w and qw in Study TDM3569g

| Dose | No. of | C <sub>max</sub> | AUCinf | T <sub>1/2</sub> | $V_d$ | CL |
|---|---|---|---|---|---|---|
| (mg/kg) | Patients | (µg/mL) | (day µg/mL) | (day) | (mL/kg) | (mL/day/kg) |
| q3w dosing | | | | | | |
| 0.3 | 3 | 9.6 (1.7) | 14.5 (3.4) | 1.3 (0.2) | 35.7 (7.5) | 21.1 (4.5) |
| 0.6 | 1 | 13.3 | 24.5 | 1.3 | 43.8 | 24.5 |
| 1.2 | 1 | 20.3 | 42.9 | 1.3 | 51.8 | 27.8 |
| 2.4 | 1 | 76.3 | 330.0 | 2.2 | 30.7 | 7.2 |
| 3.6 | 15 | 76.2 (19.1) | 300.3 (65.8) | 3.1 (0.7) | 58.4 (12.4) | 12.7 (3.6) |
| 4.8 | 3 | 130.3 (7.8) | 673.0 (12.2) | 4.1 (0.7) | 41.2 (6.2) | 7.1 (0.1) |
| qw dosing | | | | | | |
| 1.2 | 3 | 29.6 (5.7) | 76.2 (10.4) | 2.3 (0.6) | 47.5 (6.0) | 15.9 (2.4) |
| 1.6 | 3 | 34.3 (4.8) | 130.3 (39.7) | 3.4 (0.8) | 59.8 (16.6) | 13.0 (3.4) |
| 2.0 | 3 | 48.0 (9.6) | 175.0 (41.0) | 3.1 (0.3) | 51.0 (8.1) | 11.8 (2.4) |
| 2.4 | 16 | 54.8 (12.6) | 198.5 (54.5) | 3.3 (1.1) | 55.4 (13.0) | 13.1 (4.1) |
| 2.9 | 3 | 78.1 (33.9) | 212.0 (39.0) | 2.9 (0.5) | 57.7 (2.2) | 14.0 (2.6) |

AUC<sub>inf</sub> = area under the serum concentration-time curve from time 0 extrapolated to infinity;  $C_{max}$  = maximum serum concentration; CL = clearance; s.d. = standard deviation;  $T_{1/2}$  = terminal half-life;  $V_d$  = volume of distribution.

Dose intensity, defined as percentage of the planned trastuzumab emtansine dose that was actually received, was higher with the 3.6 mg/kg q3w regimen (median 99.7%, range 88%–106%) than with the 2.4 mg/kg qw schedule (median 82%, range 54%–101%). However, since the PK of trastuzumab emtansine is linear at doses  $\geq$  2.4 mg/kg, an almost 2-fold higher cumulative dose can be administered within a q3w cycle with a 2.4 mg/kg qw regimen compared with 3.6 mg/kg q3w.<sup>29,30</sup>

Based on a population PK analysis, trastuzumab emtansine has a consistent PK profile with low inter-individual variability (21%–48%) in PK parameters among patients with mBC. Greater baseline tumor burden and lower serum albumin levels, potential indicators of disease severity, resulted in small increases (< 13%) in trastuzumab emtansine clearance (CL). However, trastuzumab emtansine PK was not affected by baseline residual trastuzumab (from prior treatment) or by differences in serum concentrations of HER2 extracellular domain.<sup>35</sup>

An aggregate PK assessment of trastuzumab emtansine was performed with samples from studies TDM3569g, TDM4258g, TDM4374g, and TDM4688g. <sup>36,37</sup> PK parameters for trastuzumab emtansine, total trastuzumab, and DM1 were consistent across the four studies at Cycle 1 and steady state. Trastuzumab emtansine PK was not affected by residual trastuzumab from prior therapy or circulating extracellular domain of HER2. No significant correlations were observed between trastuzumab emtansine exposure and

efficacy, thrombocytopenia, or increased concentrations of transaminases. Across the four studies, the incidence of anti-therapeutic antibodies to trastuzumab emtansine was low and detected in 4.5% (13/286) of evaluable patients receiving trastuzumab emtansine q3w.

The PK profile (i.e., maximum concentration [ $C_{max}$ ], area under the serum concentration-time curve [AUC], terminal half-life [ $T_{1/2}$ ], apparent volume of distribution at steady state [ $V_{ss}$ ], and CL) of single-agent trastuzumab emtansine (3.6 mg/kg q3w) is predictable, well characterized, and unaffected by circulating levels of HER2 extracellular domain or residual trastuzumab. Trastuzumab emtansine exposure does not correlate with clinical responses or key AEs. Weekly administration of trastuzumab emtansine in study TDM3568g at a dose of 2.4 mg/kg showed consistent PK data with the q3w dosing schedule.<sup>29</sup>

#### 1.2.2 CAPECITABINE

Capecitabine (Xeloda<sup>®</sup>) is a fluoropyrimidine carbamate with antineoplastic activity. It is an orally administered systemic prodrug of 5'-deoxy-5-fluorouridine (5'-DFUR), which is converted to 5-fluorouracil (5-FU) in the tumor, where it inhibits DNA synthesis and slows down tumor tissue growth. It is approved in combination with docetaxel and as monotherapy in mBC. Please see the national Xeloda<sup>®</sup> prescribing information or Investigator brochure for more information.

The activity of capecitabine as single-agent chemotherapy was initially demonstrated in two multicenter Phase II clinical trials (before testing of HER2 status was standard) in patients with locally advanced or mBC after failure of a taxane and an anthracycline-containing chemotherapy regimen or for whom further anthracycline therapy was not indicated. <sup>38,39</sup> In these trials, a total of 236 patients were treated with capecitabine (1,250 mg/m² bid for 2 weeks followed by 1-week rest period). The ORRs (investigator assessment) were 20% (first trial) and 25% (second trial). The median TTP was 3.1 months and 3.2 months, respectively. Median OS was 12.6 months and 12.3 months, respectively.

The combination of capecitabine and docetaxel was studied as treatment for locally advanced or mBC after failure of anthracycline-containing chemotherapy in a multicenter randomized controlled Phase III clinical trial (SO14999). In this trial, 255 patients were randomized to treatment with capecitabine (1,250 mg/m² bid for 2 weeks followed by a 1-week rest period) and docetaxel (75 mg/m² as a 1-hour IV infusion q3w) and 256 patients were randomized to treatment with docetaxel alone (100 mg/m² as a 1-hour IV infusion q3w). OS was superior in the capecitabine plus docetaxel combination arm (HR 0.775; p = 0.0126). Median OS was 14.5 months (capecitabine plus docetaxel) *versus* 11.5 months (docetaxel alone). The ORR in the all-randomized population (investigator assessment) was 41.6% (capecitabine plus docetaxel) *versus* 29.7% (docetaxel alone; p = 0.0058). TTP was superior in the capecitabine plus docetaxel combination arm (HR 0.652; p < 0.0001). The median TTP was 6.1 months (capecitabine plus docetaxel) *versus* 4.2 months (docetaxel alone).

This trial led to the randomized Phase II CHAT trial evaluating the addition of capecitabine to first-line trastuzumab and docetaxel for locally advanced or metastatic HER2-positive mBC.<sup>41</sup> PFS was significantly improved with the addition of capecitabine (HR 0.72; median 17.9 months *versus* 12.8 months in patients receiving docetaxel and trastuzumab without capecitabine), although there was no difference in ORR (71% *versus* 73%, respectively).

### 1.2.2.1 Study BO18255: Capecitabine and Trastuzumab in LA/mGC

A global Phase III study (ToGA trial, BO18255) of trastuzumab plus chemotherapy as first-line treatment for advanced HER2-positive GC was conducted in 584 patients previously untreated for HER2-positive inoperable locally advanced or recurrent and/or metastatic adenocarcinoma of the stomach or GEJ. Patients received either capecitabine or fluorouracil combined with cisplatin or the same chemotherapy in combination with trastuzumab. The primary study endpoint was OS, defined as the time from the date of randomization to the date of death from any cause. At the time of the analysis a total of 349 randomized patients had died: 182/290 patients (62.8%) in the control arm and 167/294 patients (56.8%) in the trastuzumab-containing arm. The majority of the deaths were due to events related to the underlying cancer.<sup>18</sup>

Most patients enrolled in the study were male (76%); 52.9% were Asian and 37.7% were white. The primary tumor site was the stomach for 81.8% of patients, with the others having GEJ tumors. The addition of trastuzumab to chemotherapy resulted in an increase in median OS from 11.1 months to 13.8 months (HR 0.74, p = 0.0046). ORR (47% *versus* 35%), PFS (median 6.7 *versus* 5.5 months), and TTP (median 7.1 *versus* 5.6 months) were also significantly increased with the addition of trastuzumab to chemotherapy compared with chemotherapy alone.

With regard to OS, a treatment effect could not be excluded in any predefined subgroup, including primary tumor site, histologic subtype, method of determining HER2-positivity, performance status, chemotherapy regimen, age, gender, and region of enrollment. A multivariate analysis for OS showed a consistent result, with an adjusted HR of 0.72 (p = 0.0036); variables found to influence primary outcome included Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1 versus 2), prior gastrectomy, and Asian region of enrollment (data on file). A multivariate analysis of OS for patients enrolled in Japan, from which the bulk of Asian patients were enrolled, demonstrated a HR of 0.68. This was consistent with the overall study results.  $^{42}$ 

A pre-planned subgroup analysis by IHC score indicated that positive treatment effects were greater in tumors with higher levels of HER2 expression. Among patients whose tumors had these higher levels of HER2 expression, the median OS was 11.8 months *versus* 16 months (HR = 0.65; 95% CI: 0.51–0.83) and median PFS was 5.5 months *versus* 7.6 months (HR = 0.64; 95 % CI: 0.51–0.79) for chemotherapy *versus* chemotherapy plus trastuzumab respectively. For OS, the HR was 0.75 (95% CI: 0.51–1.11) in

the IHC 2+/FISH+ group and 0.58 (95% CI: 0.41–0.81) in the IHC 3+/FISH+ group.<sup>18</sup>

The addition of trastuzumab to chemotherapy did not result in an increased incidence of severe (Grade 3/4) or fatal AEs. There were no additional significant safety issues with trastuzumab used in the treatment of advanced GC over and above those observed when it was used in BC. Taken together, the results of the ToGA trial (BO18255) not only demonstrate the role of HER2 suppression in the treatment of HER2-positive GC but also show that HER2-directed therapies can be added to conventional chemotherapy regimens without substantial increases in side effects.

## 1.2.3 PRECLINICAL DATA OF THE COMBINATION OF TRASTUZUMAB EMTANSINE AND A FLUOROPYRIMIDINE

In preclinical BC models, additive anti-tumor activity was observed with combinations of trastuzumab emtansine and 5-FU (seeFigure 2).<sup>43</sup> In GC models a similar additive effect was observed with trastuzumab emtansine and capecitabine (see Figure 3 [data on file]).

Figure 2 MMTV HER2 Fo5 Mammary Tumor Transplants



T-DM1 = trastuzumab emtansine; 5-FU = 5-fluorouracil

Figure 3 Anti-tumor Activity of Trastuzumab Emtansine in Combination with Capecitabine in NCI-N87

T-DM1 = trastuzumab emtansine: 5-FU = 5-fluorouracil

## 1.3 STUDY RATIONALE AND RISK-BENEFIT ASSESSMENT

### 1.3.1 FOR MBC

At present, mBC remains an incurable disease. The primary goal of treatment is maximizing the patient's survival and quality of life.

HER2-positive breast tumors have been shown to benefit from anti-HER2 therapy. Regimens using the combination of anti-HER2 agents and chemotherapy have demonstrated higher efficacy than single-agent therapy. As a consequence several different combination therapies have been approved for HER2-positive mBC treatment in most countries and are considered the current standard of care.

The combination of capecitabine with anti-HER2 therapies has been shown to be beneficial in patients with HER2-positive mBC. The combination of capecitabine and lapatinib was approved in the United States in March 2007 for the treatment of patients with HER2-positive mBC who have previously received an anthracycline, a taxane, and trastuzumab. In June 2008, the European Commission granted conditional marketing authorization for lapatinib in combination with capecitabine for the treatment of patients with HER2-positive advanced or mBC whose disease has progressed on an anthracycline, a taxane, and trastuzumab in the metastatic setting. The combination of capecitabine and trastuzumab has demonstrated significant efficacy benefit when compared with capecitabine alone.

The Phase III, TDM4370g trial met its co-primary endpoint of improving PFS (by independent review) and OS compared with the combination of lapatinib and capecitabine (see Section 1.2.1.6).

Based on the studies mentioned above, the combination of trastuzumab emtansine and capecitabine could provide the potential for enhanced antitumor efficacy in mBC compared with single-agent trastuzumab emtansine or trastuzumab in combination with chemotherapy. Furthermore, preclinical data suggest that the combination of trastuzumab emtansine and capecitabine has an additive effect (see Section 1.2.3).

Approximately 2,000 patients with BC have been treated in trastuzumab emtansine clinical trials with an acceptable safety profile and a positive risk-benefit ratio. A broad development program is in place to seek approval for indications for mBC. Capecitabine in combination with an anti-HER2 agent is a proven efficacious regimen with a well-established safety profile in mBC. Trastuzumab emtansine and capecitabine have no known significant overlapping toxicities. As part of the Phase I conduct, regular teleconference calls with the investigators will be held to discuss the study treatment risk-benefit profile for each patient. An Independent Data Monitoring Committee (IDMC) will be established with the main responsibility of assessing the risk-benefit for the Phase II part of the study. Therefore, exploring the benefit of combination therapy of trastuzumab emtansine and capecitabine in patients with mBC seems justified.

## 1.3.2 FOR MGC

As for mBC, the primary goal of treatment for metastatic gastric cancer (mGC) is to maximize patients' survival and quality of life.

In HER2-positive gastric tumors, anti-HER2 therapy has shown benefit. In the ToGA study (BO18255), the combination of chemotherapy and trastuzumab significantly improved OS versus chemotherapy alone (see Section 1.2.2.1) in this population. Fluoropyrimidine-based therapies (capecitabine, 5-FU) are the standard of care in mGC in general and were also the most frequent combination agents used in the ToGA trial (BO18255; see Section 1.2.2.1).

Furthermore, preclinical data suggest that the combination of trastuzumab emtansine and capecitabine has an additive effect (see Section 1.2.3).

A development program for trastuzumab emtansine is in place to seek approval for mGC indications. Capecitabine in combination with trastuzumab is a proven efficacious regimen with a well-established safety profile in mGC. Trastuzumab emtansine and capecitabine might have overlapping toxicities and therefore safety monitoring is in place to avoid exposing patients to harm. Therefore, exploring the benefit of combination therapy of trastuzumab emtansine and capecitabine in patients with mGC seems justified.

In the ToGA study in LA/mGC, trastuzumab exposure was lower than that observed in breast cancer studies. Based on this observation, together with pharmacokinetic results and findings from a Phase I study in mBC, it was considered that a weekly trastuzumab emtansine regimen may provide higher

cumulative trastuzumab emtansine exposure than the q3w schedule and was therefore chosen for the Phase I, Cohort 2 part of the present study in LA/mGC. This approach has subsequently been supported by findings from stage I of the adaptive phase II/III BO27952 trial in this setting (see Section 3.3.2.2). In October 2013, the IDMC for the BO27952 trial recommended selection of the weekly 2.4 mg/kg regimen for further evaluation in the phase III part of the trial based on pharmacokinetic, safety, and efficacy data available at the time.

Results from the Phase I part of the study in mGC will be used as supporting information for future studies in the indication.

## 2. OBJECTIVES

## 2.1 PHASE I: MTD-FINDING OF TRASTUZUMAB EMTANSINE AND CAPECITABINE IN MBC

### 2.1.1 PRIMARY OBJECTIVE

 To determine the MTD of the combination of trastuzumab emtansine and capecitabine in patients with HER2-positive mBC

#### 2.1.2 SECONDARY OBJECTIVES

To assess the:

- PK of trastuzumab emtansine, capecitabine and their metabolites
- Safety of the combination of trastuzumab emtansine and capecitabine
- ORR

# 2.2 RANDOMIZED PHASE II: EXPLORATION OF EFFICACY AND SAFETY IN MBC

#### 2.2.1 PRIMARY OBJECTIVE

To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone in patients with HER2-positive mBC, as measured by ORR by RECIST v.1.1 per investigator local assessment

#### 2.2.2 SECONDARY OBJECTIVES

To assess the safety profile of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone

To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone in patients with HER2-positive mBC, as measured by:

- Time to response (TTR)
- DoR

- TTP
- TTF
- PFS
- CBR
- OS

## 2.3 PHASE I: MTD FINDING OF TRASTUZUMAB EMTANSINE AND CAPECITABINE IN LA/MGC

#### 2.3.1 PRIMARY OBJECTIVE

To determine the MTD of the combination of trastuzumab emtansine and capecitabine in patients with LA/mGC

#### 2.3.2 SECONDARY OBJECTIVES

To assess the:

- PK of trastuzumab emtansine, capecitabine, and their metabolites
- Safety of the combination of trastuzumab emtansine and capecitabine
- ORR

## 3. <u>STUDY DESIGN</u>

### 3.1 DESCRIPTION OF STUDY

This is an international, multicenter Phase I/II dose-finding study of two dosing schedules of trastuzumab emtansine and capecitabine combination therapy in HER2-positive mBC and LA/mGC.

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in Phase I studies in patients with HER2-positive mBC or LA/mGC.

The efficacy and safety of the combination in patients with mBC will also be explored in a randomized, open-label Phase II part of the study.

## 3.1.1 OVERVIEW OF STUDY DESIGN

### **Overview of Study Design**

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with HER2-positive mBC or LA/mGC using a Phase I design, followed by a randomized, open-label Phase II part of the study to explore the efficacy and safety of the combination in patients with HER2-positive mBC. There will be no follow-on randomized exploration of efficacy in mGC. Results from the Phase I study in LA/mGC will be used as supporting information for future studies in the indication.

Cohort 1 for patients with mBC will open first and the MTD will be established. Once the MTD is defined, both the randomized Phase II trial for patients with
HER2-positive mBC and the Phase I Cohort 2 for patients with LA/mGC will open.

An overview of the study design is depicted in Figure 4.

# **Duration of Treatment and Patient Follow-up**

<u>Duration of treatment:</u> All patients will be treated until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor. If toxicity is considered by the investigator to be related to only one of the two agents, the non-implicated agent can be continued as single-agent therapy.

If at the time of study closure there are patients whose disease has not progressed and who are still receiving study treatment, they will be offered the possibility to continue treatment by enrolling in an extension study at the discretion of the investigator.

<u>Patient follow-up:</u> All patients will be followed up until withdrawal of consent, death, or for up to a maximum of 2 years after the last patient was randomized in the Randomized Phase II part of the study, whichever occurs first.

# **Duration of Study, Database Closure and Data Reporting**

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to last 2 years in total (1 year for the MTD-Finding study in mBC and 1 year for the Phase II Exploration of Efficacy and Safety in mBC). See Section 3.2 for further details about EOS.

Specifically in Phase I, cohort 2, if dose level -2 is too toxic in LA/mGC, recruitment into the LA/mGC cohort will be closed. See Section 3.1.1.3 for details of treatment continuation if patients are still responding to treatment at this time.

Data may be published/presented publicly at the end of each cohort e.g., once the MTD for Cohort 1 for mBC has been defined and the dose for Phase II Exploration of Efficacy and Safety has been selected, and after the prespecified analyses for the Randomized Phase II exploration of efficacy and safety in mBC. The Clinical Study Report (CSR) will be finalized/published within 1 year after EOS (LPLV).

Figure 4 Overview of Study Design



<sup>&</sup>lt;sup>1</sup> Capecitabine doses are administered daily on Days 1–14 q3w

mBC = metastatic breast cancer; LA/mGC = locally advanced/metastatic gastric cancer; MTD = maximum tolerated dose; q3w = every 3 weeks; qw = weekly.

A schedule of assessments is provided in Appendix 1.

# 3.1.1.1 Overview of Phase I Design in Patients with mBC

An overview of the Phase I study design is depicted in Figure 5.

<sup>&</sup>lt;sup>2</sup> The MTD defined in the mBC Phase I study will be implemented in the mBC Randomized Phase II and mGC Phase I studies

<sup>&</sup>lt;sup>3</sup> Cohort 2 will open to recruit patients with LA/mGC using the MTD defined in Phase I for patients with mBC. Dose Level 1 will not be explored in Cohort 2 (see also Section 3.3.2.2)

<sup>&</sup>lt;sup>4</sup> Stratification factor: Number of prior lines of treatment for metastatic disease (≤1 or >1; excluding single-agent hormones)



Figure 5 Overview of Phase I Dose Finding Study Design

DLT = dose-limiting toxicity; MTD = maximum tolerated dose

## Determination of the MTD in Patients with mBC

The trial will first investigate the feasibility of the combination of capecitabine and trastuzumab emtansine q3w in one cohort of up to 18 patients, by deescalating the dose of capecitabine from 750 mg/m² bid to 650 mg/m² bid on Days 1 to 14 q3w with a 3 plus 3 classical Phase I design. Cohort 1 will open first and enroll patients with HER2-positive mBC.

#### **Enrollment into Cohort 1**

# MTD-finding in patients with mBC (Phase I)

According to the 3 plus 3 classical study design, Cohort 1 will start with the enrollment of 3 patients at Dose Level 1. Patients will be evaluated for DLTs as specified in the DLT definition (see Section 5.1.4). The dose of trastuzumab emtansine is fixed at 3.6 mg/kg q3w. Three dose levels of capecitabine administered bid on Days 1 to 14 q3w will be tested.

The following doses will be explored in Cohort 1:

**Dose Level 1:** 750 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine

<sup>&</sup>lt;sup>1</sup>Repeat with the new dose level until the MTD is established

<sup>&</sup>lt;sup>2</sup> If Dose Level -2 is too toxic (DLT in > 1/6 patients), the study will be terminated.

**Dose Level -1:** 700 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine

**Dose Level -2:** 650 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine

The following MTD determining rules will be applied during the MTD-Finding treatment phase:

- Step 1: Three patients will be enrolled at Dose Level 1
- Step 2: The toxicity of Dose Level 1 will be monitored and the following actions taken:
  - a) If none of these 3 patients (0/3) experiences a DLT, the MTD will be established as the current dose level and will need to be confirmed in 3 more patients (to achieve DLTs in ≤ 1/6 patients at that dose level)
  - b) If 1 of the initial 3 patients (1/3) experiences a DLT, an additional 3 patients should be enrolled and treated at the same dose, i.e., Dose Level 1
  - c) If no additional patients experience a DLT (1/6), the MTD will be established as the current dose level
  - d) If 1 or more additional patients experience a DLT (> 1/6), the dose will be de-escalated to the next lowest dose level. If no more than 1 patient experiences a DLT (≤ 1/6) after dose de-escalation, the dose will be considered the MTD and, following IDMC recommendation, will be further explored in the Randomized Phase II part of the study. Dose re-escalation will not be allowed. If 2 or more patients experience a DLT (> 1/6) after dose de-escalation, de-escalation should continue to the next lowest dose level. Based on the DLT findings, the next dose level may be considered the MTD and, following IDMC recommendation, be further explored in the Randomized Phase II part of the study or the study may be terminated if DLTs occur in > 1/6 patients at Dose Level -2.

In order to define the dose for the Randomized Phase II Exploration of Efficacy and Safety part of the study, evaluation will include not only the DLTs during Cycle 1 but also all available safety information during the subsequent cycles. The dose level considered optimal will be the dose level selected to proceed to the Phase II and LA/mGC parts of the study.

Once the appropriate dose of study medication is established, the Randomized Phase II part of the study and Phase I, Cohort 2 will open as shown in Figure 4.

# 3.1.1.2 Overview of Phase II: Exploration of Efficacy and Safety in Patients with mBC

After review of safety data from Part 1, cohort 1, the IDMC recommended a regimen of capecitabine 700 mg/m<sup>2</sup> bid days 1–14 in combination with trastuzumab emtansine 3.6 mg/kg q3w for further evaluation. The Phase II part of the study will explore the efficacy and safety of this recommended

regimen compared with trastuzumab emtansine alone in patients with HER2-positive mBC. See Section 3.1.1 for details of duration of treatment.

Approximately 210 additional patients with HER2-positive mBC will be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to the Phase II part of the study; however, they will be followed-up until end of study (EOS).

# 3.1.1.3 Overview of Phase I Design in LA/mGC Patients

#### Determination of the MTD in Patients with LA/mGC

Cohort 2 will enroll patients with HER2-positive LA/mGC. Trastuzumab emtansine will be administered qw at a fixed dose of 2.4 mg/kg and capecitabine will be started at 700 mg/m<sup>2</sup> bid, the MTD defined for patients with mBC in Cohort 1.

#### **Enrollment into Cohort 2**

Cohort 2 will open with a 3 plus 3 classical design to investigate the feasibility of combination therapy of capecitabine and trastuzumab emtansine in up to 12 patients with LA/mGC. The capecitabine dose will be de-escalated from the starting dose of 700 mg/m² bid (the MTD recommended in Cohort 1).

The dose levels for de-escalation of capecitabine will be the same as described for Cohort 1, except for Dose Level 1, which will not be explored in patients with mGC (see also Section 3.3.2.2).

If Dose Level -1 (700 mg/m<sup>2</sup> bid, the MTD recommended in cohort 1) is well tolerated (DLT in  $\leq$  1/6), this dose will be established as the MTD for LA/mGC.

- If Dose Level -1 is not tolerated in Cohort 2 (DLT in > 1/3 or > 1/6 patients), de-escalation will be to Dose Level -2.
- If Dose Level -2 is not tolerated in Cohort 2 (DLT in > 1/6), the combination will be considered not feasible in LA/mGC and Cohort 2 will be terminated. Patients who, at that time, experience response according to RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the Steering Committee (SC).

#### 3.1.1.4 Number of Patients

Overall, it is anticipated that the maximum number of patients enrolled into the study will be approximately 240.

# Phase I, Cohort 1: mBC

Between 6 and 18 patients will be enrolled into Cohort 1 to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with mBC.

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

For this part of the study, a total of approximately 210 patients with mBC will be randomized.

# Phase I, Cohort 2: mGC

After the MTD in Cohort 1 has been established, 3–12 patients will be enrolled into Cohort 2 to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with mGC.

#### 3.1.1.5 Number of Centers

This is a multicenter, international study.

## 3.1.2 STEERING COMMITTEE

A SC has been established for this study. Initially, it is composed of the investigators participating in the Phase I, Cohort 1 part of the study and one medical representative and one statistician of the Sponsor. The study design and DLT definition have been developed by the SC. See the SC Charter for further information.

The SC will collectively review the status of the ongoing patients in Phase I on a regular basis. The SC will adjudicate in the event of DLTs that are not covered by the existing DLT criteria.

## 3.1.3 INDEPENDENT DATA MONITORING COMMITTEE

An IDMC will review the safety outcomes for patients enrolled in Phase I, Cohort 1 and recommend whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 25, 75, and 150 patients have received at least 3 cycles (Cycle 3 Day 21) of treatment in the Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II part of the study or as requested.

# 3.2 END OF STUDY

EOS is defined as the last patient last visit (LPLV) at the end of the follow-up period, as defined in Section 3.1.1. This will be the last data collection point, which can be a clinic visit or a laboratory sample. LPLV is expected to occur approximately 2 years after the last patient has been randomized into the Phase II part of the trial.

## 3.3 RATIONALE FOR STUDY DESIGN

## 3.3.1 RATIONALE FOR PATIENT GROUP SELECTION

Nonclinical studies indicate that the sensitivity of cancer cells to trastuzumab emtansine requires HER2 overexpression, and measurement of such expression is a standard of care in determining eligibility for trastuzumab therapy (see the Herceptin® national prescribing information). Measurement of

HER2 gene amplification has traditionally been performed using IHC. HER2 gene amplification determined by ISH has also proven to be a reliable method for demonstrating HER2-positive status.<sup>44</sup>

This study will enroll patients diagnosed with HER2-positive mBC or LA/mGC. Capecitabine is an established chemotherapy for both diseases. In patients with HER2-positive mBC or LA/mGC, anti-HER2 therapy has demonstrated activity. Furthermore, the combination of anti-HER2 therapy and capecitabine has been shown to be efficacious in both mBC<sup>9,10</sup> and LA/mGC.<sup>18</sup> Eligible patients for this study will have incurable mBC or LA/mGC overexpressing HER2.

## 3.3.1.1 Rationale for Phase I

The 3 plus 3 design is a well-established and well-known method for Phase I studies. PK parameters will be collected and analyzed to investigate the PK interaction of the drugs under investigation.

The capecitabine dose evaluated in combination with trastuzumab and docetaxel in the CHAT trial was 950 mg/m² bid. However, retrospective evaluations and post hoc analyses of early dose reduction suggest that lower starting doses of capecitabine offer similar efficacy with better tolerability. Therefore the capecitabine starting dose selected in combination with trastuzumab emtansine for the MTD-Finding Phase I part of the present study was 750 mg/m² bid, taking into account the aim of maintaining the good tolerability of trastuzumab emtansine while benefitting from synergy observed between the two agents in nonclinical studies.

The combination of T-DM1 and capecitabine was evaluated with a deescalation study design. Following the emergence of two DLTs (grade 3 vomiting, grade 3 elevated AST/ALT) at the starting dose of 750 mg/m² bid (days 1–14 q3w) in combination with trastuzumab emtansine 3.6 mg/kg q3w, a de-escalated dose cohort was opened to evaluate capecitabine 700 mg/m² bid combined with the same dose of trastuzumab emtansine. At this dose no DLTs were observed in the six patients treated, and of note, none of the patients had experienced grade ≥3 AEs in cycles delivered after the DLT evaluation period.<sup>45</sup> Following review of safety data from patients treated at these two dose levels, the IDMC recommended the regimen of capecitabine 700 mg/m² bid combined with trastuzumab emtansine 3.6 mg/kg q3w for the phase II exploration of efficacy and safety.

In the ToGA study in LA/mGC, trastuzumab exposure was lower than that observed in breast cancer studies. A weekly trastuzumab emtansine regimen may provide higher cumulative trastuzumab emtansine exposure than the q3w schedule and was therefore chosen for the Phase I, Cohort 2 part of the present study in LA/mGC. This approach has subsequently been supported by findings from stage I of the adaptive phase II/III BO27952 trial in this setting (see Section 3.3.2.2).

#### 3.3.1.2 Rationale for Randomized Phase II

The Randomized Phase II part of the study is designed to explore the efficacy and safety of the combination recommended following the Phase I MTD-Finding phase (trastuzumab emtansine 3.6 mg/kg in combination with capecitabine 700 mg/m²) compared with trastuzumab emtansine alone.

# 3.3.2 RATIONALE FOR INVESTIGATIONAL MEDICINAL DOSE SELECTION

## 3.3.2.1 In Patients with mBC

In study TDM3569g, the MTD of trastuzumab emtansine administered by IV infusion q3w was 3.6 mg/kg. As described in Section 1.2, clinical activity has been observed at a dose of 3.6 mg/kg q3w in two Phase II studies of single-agent trastuzumab emtansine in patients with heavily pre-treated HER2-positive mBC (protocol TDM4258g<sup>31</sup> and protocol TDM4374g<sup>32</sup>), in patients who had not received prior chemotherapy for metastatic disease (TDM4450g<sup>26</sup>), and subsequently in the randomized phase III trials.<sup>27,28</sup>

Capecitabine doses have been selected as being in the range of efficacious doses for single-agent or combination use. The doses selected are within the dosing range included in the Xeloda® Summary of Product Characteristics (SmPC) and therefore are considered to be efficacious.

#### 3.3.2.2 In Patients with mGC

In the ToGA study (BO18255) evaluating trastuzumab in combination with chemotherapy for mGC, patients with higher drug exposure had a greater benefit than those with lower exposure.<sup>46</sup> As a consequence, an ongoing randomized, open-label, multicenter Phase IIIb study is comparing two trastuzumab dosing regimens, each in combination with cisplatin/capecitabine chemotherapy, as first-line therapy in patients with HER2-positive metastatic gastric or GEJ adenocarcinoma (Study BO27798).

In TDM3569g (see Section 1.2.1.1), the qw administration of 2.4 mg/kg of trastuzumab emtansine resulted in higher exposure than q3w dosing (see Section 1.2.1.8).<sup>29,30</sup> Therefore, this dose may result in larger clinical benefit for patients with mGC.

In the ongoing randomized adaptive phase II/III BO27952 trial evaluating trastuzumab emtansine versus the investigator's choice of taxane therapy in unrectable LA/mGC, two trastuzumab emtansine regimens were evaluated in stage I: 3.6 mg/kg q3w and 2.4 mg/kg qw . In October 2013, the IDMC for the BO27952 trial recommended selection of the weekly 2.4 mg/kg regimen for further evaluation in the phase III part of the trial based on pharmacokinetic, safety, and efficacy data available at the time. This recommendation provides further support for using the weekly regimen in Phase I, Cohort 2 of the present trial.

In Cohort 2, the starting dose of capecitabine will be 700 mg/m<sup>2</sup> bid (the MTD from Cohort 1 in mBC) in order to minimize the exposure of patients to suboptimal treatment. The dose of capecitabine can be de-escalated if needed.

#### 3.3.2.3 Rationale for Duration of Treatment

Treatment will be given until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor (see Section 3.1.1 for full information). As of 1 January 2010, of 237 patients enrolled in studies TDM3569g, TDM4258g, and TDM4374g receiving trastuzumab emtansine at 3.6 mg/kg, approximately 30% have tolerated more than 12 cycles, with 14.8% having received more than 17 cycles. Twenty patients (8.4%) have discontinued trastuzumab emtansine due to AEs and 24 patients (10.1%) required dose reductions in trastuzumab emtansine because of AEs. In the absence of unacceptable toxicity, patients with mBC are generally treated until PD. Further support for treatment until PD comes from the EMILIA randomized phase III trial.<sup>27</sup> Among the 490 patients randomized to trastuzumab-emtansine, only 29 (5.9%) discontinued because of adverse events.

Capecitabine will be given until PD, in accordance with Xeloda® national prescribing information.

# 3.3.3 PHARMACOKINETIC SAMPLING RATIONALE

PK is studied only in the Phase I (MTD-Finding) parts (both cohorts 1 and 2). The PK sampling rationale is to characterize the PK of trastuzumab emtansine and capecitabine and their metabolites, to assess any potential drug-drug interaction when trastuzumab emtansine is given in combination with capecitabine, and to explore potential correlations between drug exposure and measures of both efficacy (ORR) and toxicity (alanine transaminase [ALT]/AST, platelets, etc.), if data allow.

## 3.4 OUTCOME MEASURES

## 3.4.1 PHASE I: MBC

# 3.4.1.1 Primary Outcome Measure

The main objective for Phase I is to determine the MTD of capecitabine when combined with trastuzumab emtansine.

## 3.4.1.2 Secondary Outcome Measure

The secondary outcome is ORR, based on best overall response (BOR) rate according to RECIST v.1.1, per investigator local assessment.

# 3.4.1.3 Primary Safety Outcome Measure

The primary safety outcome measure is to establish the MTD. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination and will be summarized for each treatment dosage.

# 3.4.1.4 Secondary Safety Outcome Measures

Safety endpoints will be summarized for each treatment dosage:

- Incidence, nature, and severity of AEs, according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v. 4.0
- Incidence, nature, and severity of SAEs, according to NCI CTCAE v. 4.0
- Incidence and nature of Grade ≥3 AEs
- Incidence, nature, and severity of AEs of special interest (AESIs), according to NCI CTCAE v. 4.0
- Fatal AEs and their causes
- Laboratory parameters
- LVEF
- Exposure to study medication
- Physical examination
- Vital signs and ECOG performance status
- Premature withdrawal from study medication and/or study

#### 3.4.1.5 Pharmacokinetic Outcome Measures

The PK outcome measures to be assessed in patients receiving trastuzumab emtansine and capecitabine will include:

- Serum concentrations of trastuzumab emtansine (conjugated drug) and total trastuzumab (free and conjugated to DM1)
- Plasma concentration of DM1
- Plasma concentration of capecitabine and its active metabolite 5-FU
- Total exposure (e.g., AUC)
- Cmax
- CL
- V<sub>d</sub>
- T<sub>1/2</sub>

# 3.4.2 RANDOMIZED PHASE II: EXPLORATION OF EFFICACY AND SAFETY IN MBC

The primary and secondary efficacy outcome measures will be presented for each treatment group.

# 3.4.2.1 Primary Efficacy Outcome Measure

The primary outcome measure is ORR by investigator assessment, based on BOR (defined as the best response recorded from randomization into the Phase II part of the study and until PD, death, withdrawal of consent, start of

new anticancer treatment, or EOS, whichever occurs first) according to RECIST v.1.1 (See Appendix 3).

# 3.4.2.2 Secondary Efficacy Outcome Measures

Secondary efficacy outcomes include:

- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

# 3.4.2.3 Primary Safety Outcome Measure

A primary safety outcome is defined only for Phase I.

# 3.4.2.4 Secondary Safety Outcome Measures

The summary of safety endpoints will be presented for each treatment group:

- Incidence, nature, and severity of AEs, according to NCI CTCAE v. 4.0
- Incidence, nature, and severity of SAEs, according to NCI CTCAE v. 4.0
- Incidence and nature of Grade ≥3 AEs
- Incidence, nature, and severity of AESIs, according to NCI CTCAE v. 4.0
- Fatal AEs and their causes
- Events to monitor
- Laboratory parameters
- LVEF
- Exposure to study medication
- Physical examination
- Vital signs and ECOG performance status
- Premature withdrawal from study medication and/or study

# 3.4.2.5 Pharmacokinetic Outcome Measures

Not applicable for Phase II.

## 3.4.3 Phase I: LA/MGC

# 3.4.3.1 Primary Outcome Measure

The main objective for Phase I is to determine the MTD of capecitabine when combined with trastuzumab emtansine. The number and the proportion of

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 3, 30 June 2014

55

patients with DLTs will be used as the primary measure for the MTD determination and will be summarized for each treatment dosage.

# 3.4.3.2 Secondary Efficacy Outcome Measure

The secondary (efficacy) outcome is ORR, based on BOR rate according to RECIST v.1.1 according to investigator assessment.

## 3.4.3.3 Secondary Safety Outcome Measures

Safety endpoints will be summarized for each treatment dosage:

- Incidence, nature, and severity of AEs, according to NCI CTCAE v. 4.0
- Incidence, nature, and severity of SAEs, according to NCI CTCAE v. 4.0
- Incidence and nature of Grade ≥3 AEs
- Incidence, nature, and severity of AESIs, according to NCI CTCAE v. 4.0
- Fatal AEs and their causes
- Events to monitor
- Laboratory parameters
- LVEF
- Exposure to study medication
- Physical examination
- Vital signs and ECOG performance status
- Premature withdrawal from study medication and/or study

# 3.4.3.4 Pharmacokinetic Outcome Measures

The PK outcome measures to be assessed in patients receiving trastuzumab emtansine and capecitabine will include:

- Serum concentrations of trastuzumab emtansine (conjugated drug) and total trastuzumab (free and conjugated to DM1)
- Plasma concentration of DM1
- Plasma concentration of capecitabine and its active metabolite 5-FU
- Total exposure (e.g., AUC)
- Cmax
- CL
- V<sub>d</sub>
- T<sub>1/2</sub>

# 4. MATERIALS AND METHODS

# 4.1 PATIENTS

## 4.1.1 PATIENTS WITH MBC

This study will enroll patients with HER2-positive BC with histologically or cytologically confirmed metastatic disease that is amenable to combination treatment with trastuzumab emtansine and capecitabine.

Patients with mBC must have received at least one prior treatment regimen for early or metastatic disease, which included a chemotherapy agent and trastuzumab either separately or in combination. In both study parts (Phase I and II), only patients whose HER2 tumor status was locally scored as IHC 3+ or in situ hybridization (ISH) positive will be eligible.

# 4.1.2 LA/MGC PATIENTS

This study will enroll patients with HER2-positive GC with histologically or cytologically confirmed inoperable LA/mGC that is amenable to combination treatment with trastuzumab emtansine and capecitabine.

Patients with mGC must not have received prior chemotherapy for advanced/metastatic disease, and only patients with HER2-positive primary tumor or metastasis as assessed by the central laboratory will be allowed to enroll in the mGC part of the study.

## 4.1.3 INCLUSION CRITERIA

#### 4.1.3.1 For Patients with mBC

Patients must meet the following criteria for study entry:

- 1. Male or female
- 2. Age ≥ 18 years old
- 3. Signed informed consent before any study-specific procedure
- 4. Able and willing to comply with the protocol
- 5. Negative serum pregnancy test for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in the medical history confirming that the patient is not of childbearing potential.
- 6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 7 months after the last dose of study treatment (see Section 5.2.4).

- 7. ECOG performance status of 0, 1, or 2
- 8. Blood:
  - a) Platelet count > 100,000 cells/mm<sup>3</sup>
  - b) International normalized ratio (INR) < 1.5
  - c) Absolute neutrophil count (ANC) > 1,500 cells/mm<sup>3</sup>
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 9. Liver function:
  - a) Total bilirubin ≤ 1.5 × upper limit of normal (ULN) or direct bilirubin ≤1.5 × ULN in patients with documented Gilbert's syndrome.
  - b) Serum glutamic oxaloacetic transaminase (SGOT)/AST and serum glutamic pyruvic transaminase (SGPT)/ALT ≤ 2.5 × ULN
  - c) Alkaline phosphatase  $\leq 2.5 \times ULN$ . In patients with bone metastases: alkaline phosphatase  $\leq 5 \times ULN$
  - d) Evidence of stable liver function during the month prior to enrollment with liver function test (LFT) fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin).
- 10. Renal function:
  - a) Serum creatinine of < 177 µmol/L or calculated creatinine CL > 50 mL/min. If urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate ≤ 1 g of protein/24 hours
- 11. Cardiac function:
  - a) LVEF ≥ 50% by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan
- 12. Life expectancy ≥12 weeks
- 13. Histologically or cytologically confirmed BC
- 14. HER2-positive disease, defined as IHC 3+ or ISH positive
- 15. Tumor block or 8 slides available for retrospective central confirmation of HER2-positivity (central confirmation not necessary for enrollment).
- 16. mBC with at least one measurable lesion according to RECIST v.1.1
- 17. Disease progression on at least one prior regimen containing trastuzumab and chemotherapy either separately or in combination
- 18. Patients must have recovered from previous treatments

## 4.1.3.2 For Patients with LA/mGC

Patients must meet the following criteria for study entry:

- 1. Male or female
- 2. Age ≥ 18 years old
- 3. Signed informed consent before any study-specific procedure

- 4. Able and willing to comply with the protocol
- 5. Negative serum pregnancy test for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in the medical history confirming that the patient is not of childbearing potential
- 6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 7 months after the last dose of study treatment (see Section 5.2.4)
- 7. ECOG performance status of 0, 1, or 2
- 8. Blood:
  - a) Platelet count > 100,000 cells/mm<sup>3</sup>
  - b) INR < 1.5
  - c) ANC > 1,500 cells/mm<sup>3</sup>
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 9. Liver function:
  - a) Total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤1.5 × ULN in patients with documented Gilbert's syndrome
  - b) SGOT/AST and SGPT/ALT ≤ 2.5 × ULN
  - c) Alkaline phosphatase ≤ 2.5 × ULN. In patients with bone metastases: alkaline phosphatase ≤ 5 × ULN
  - d) Evidence of stable liver function in the month prior to enrollment with LFT fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin).
- 10. Renal function:
  - a) Serum creatinine of < 177 µmol/L or calculated creatinine CL > 50 mL/min. If urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate ≤ 1 g of protein/24 hours
- 11. Cardiac function:
  - a) LVEF ≥ 50% by ECHO or MUGA scan
- 12. Histologically or cytologically confirmed mGC or locally advanced GC
- 13. HER2-positive tumor (primary tumor or metastatic lesion), defined as either IHC 3+ or IHC 2+ and ISH+, prospectively confirmed by a Sponsor-designated central laboratory prior to enrollment. ISH positivity is defined

as a ratio of  $\geq$  2.0 for the number of HER2 gene copies to the number of signals for CEP17.

- a) Archival tumor samples obtained from primary or metastatic sites are acceptable.
- b) Invasive tumor for central confirmation of HER2 status is required.
- c) A formalin-fixed paraffin-embedded (FFPE) tissue block with at least 5 mm of invasive tumor for central confirmation is preferred. If FFPE tissue blocks (or partial block) are unavailable due to country or site regulations, a minimum of 8 freshly cut unstained slides MUST be available for central review of HER2 status.
- 14. Inoperable LA/mGC

## 4.1.4 EXCLUSION CRITERIA

#### 4.1.4.1 For Patients with mBC

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half-lives, whichever is longer
  - b) Hormonal therapy within 14 days
  - c) Trastuzumab within 21 days
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine
- 3. Prior treatment with capecitabine
- 4. History of severe and unexpected reactions to fluoropyrimidine or known hypersensitivity to fluorouracil
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogues, such as brivudine
  - b) Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
  - c) Signs or symptoms suggesting that the patient has DPD deficiency
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>
  - b) Epirubicin > 900 mg/m<sup>2</sup>
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m<sup>2</sup> doxorubicin.

- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 28 days before first study drug administration
- Current peripheral neuropathy of Grade ≥ 3 according to NCI CTCAE, v. 4.0
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above.
- 11. Current unstable ventricular arrhythmia requiring treatment
- 12. History of symptomatic CHF (New York Heart Association [NYHA] Classes II–IV)
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
- 15. Severe dyspnea at rest due to complications of advanced malignancy or currently requiring continuous oxygen therapy
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation
- 20. Current known active infection with human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C virus (HBV/HCV)
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Lapatinib ≤ 14 days before first study drug administration
- 22. Previous radiotherapy for the treatment of mBC is not allowed if:
  - a) The last fraction of radiotherapy has been administered within 14 days prior to first study drug administration (28 days for patients with radiotherapy to control symptoms of brain metastases, see exclusion criterion 8).
  - b) More than 25% of marrow-bearing bone has been irradiated.
  - c) Any acute toxicity has not resolved to Grade ≤ 1 before first study drug administration

#### 4.1.4.2 For Patients with LA/mGC

- Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half-lives, whichever is longer
  - b) Hormonal therapy within 14 days
  - c) Trastuzumab within 21 days
- 2. Prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received prior trastuzumab emtansine
- 3. Prior treatment with capecitabine
- 4. History of severe or unexpected reactions to fluoropyrimidine or known hypersensitivity to fluorouracil
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogs, such as brivudine
  - b) Rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
  - c) Signs or symptoms suggesting that the patient has DPD deficiency
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>
  - b) Epirubicin > 900 mg/m<sup>2</sup>
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control symptoms within 28 days before first study drug administration
- Current peripheral neuropathy of Grade ≥ 3 according to NCI CTCAE, v. 4.0
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above
- 11. Current unstable ventricular arrhythmia requiring treatment
- 12. History of symptomatic CHF (NYHA Classes II-IV)
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration

- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
- 15. Severe dyspnea at rest due to complications of advanced malignancy or currently requiring continuous oxygen therapy
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation
- 20. Current known active infection with HIV, HBV, and/or HCV
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Previous chemotherapy for advanced/metastatic disease
  - a) Prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrollment into the study
- 22. Lapatinib ≤ 14 days before first study drug administration

#### 4.1.5 PATIENT REPLACEMENT POLICY

None of the patients in the Phase I part of the study may be replaced unless approved by the entire SC. Phase II patients will not be replaced.

### 4.2 METHOD OF TREATMENT ASSIGNMENT

In the Randomized Phase II part of the study, patients will be randomized to receive either the combination of trastuzumab emtansine and capecitabine or trastuzumab emtansine alone. Patients are stratified according to the number of prior lines of treatment for metastatic disease (≤1 or >1, excluding single-agent therapy).

This is an open-label randomized study; therefore, no blinding will be used.

# 4.3 STUDY TREATMENT

# 4.3.1 FORMULATION, PACKAGING, AND HANDLING

## 4.3.1.1 Trastuzumab Emtansine

Trastuzumab emtansine is provided as a single-use, lyophilized formulation in a colorless 20 mL Type I glass vial containing 160 mg of trastuzumab emtansine, closed by means of a FluroTec coated stopper and an overseal with flip-off cap. Upon receipt of trastuzumab emtansine, vials should be

refrigerated at 2–8°C (36–46°F) until use. THE VIAL MUST NOT BE FROZEN OR SHAKEN. Trastuzumab emtansine must be stored in the original carton to protect it from light. Do not use the product beyond the expiration date provided by the manufacturer. Any remaining medication should be discarded.

All vials of trastuzumab emtansine should be handled by appropriately trained site staff wearing gloves and using appropriate procedures in place at the clinical site for preparation of chemotherapeutic drugs. Vials should be visually inspected upon receipt to ensure that they are intact without exterior contamination. Discard any cracked vials and report vials with surface contamination to the clinical site manager for assessment.

The lyophilized product should be reconstituted using sterile water for injection (SWFI). Using a new syringe, 8 mL SWFI should be added to the vial and the vial swirled gently until the product is completely dissolved. The vial should not be shaken. The resulting product contains 20 mg/mL trastuzumab emtansine, 10 mM sodium succinate, pH 5.0, 60 mg/mL sucrose, and 0.02% (w/v) polysorbate 20. Each 20 mL vial contains enough trastuzumab emtansine to allow delivery of 160 mg trastuzumab emtansine. The reconstituted product contains no preservative and is intended for single use only.

The vial should be inspected to ensure the reconstituted product is a clear colorless solution, and is free of particulates before proceeding. Drug from any vial that appears abnormal upon inspection should not be administered to patients. Using a new syringe, the indicated volume of trastuzumab emtansine solution should be removed from the vial(s) and added to the IV bag containing at least 250 mL of 0.45% sodium chloride (preferred) or 0.9% sodium chloride injection and gently inverted to mix the solution. A 0.22 micron non-protein adsorptive polyethersulfone in line filter is recommended when using 0.45% sodium chloride and required when using 0.9% sodium chloride injection. The solution of trastuzumab emtansine should not be shaken.

The solution of trastuzumab emtansine for infusion should be used immediately. If not used immediately, storage times should not be longer than 24 hours at 2–8°C (36–46°F) for solutions of trastuzumab emtansine diluted in polyvinyl chloride (PVC) or latex free PVC-free polyolefin, polypropylene, or polyethylene bags containing 0.45% or 0.9% Sodium Chloride for Injection.

For additional details, please refer to the current version of the trastuzumab emtansine Investigator's Brochure.

# 4.3.1.2 Capecitabine

The following information has been obtained from the Xeloda® European Union (EU) SmPC and US Xeloda® Package Insert.

Capecitabine is available as biconvex, oblong, film-coated tablets, available as follows:

• 150 mg tablets: color, light peach; engraving, XELODA on one side, 150 on the other; packs of 60

• 500 mg tablets: color, peach; engraving, XELODA on one side, 500 on the other; packs of 120

Capecitabine tablets should not be stored above 30°C.

## 4.3.2 DOSAGE AND ADMINISTRATION

#### 4.3.2.1 For Patients with mBC

#### **Trastuzumab Emtansine**

Trastuzumab emtansine will be administered on Day 1 q3w at a dose of 3.6 mg/kg IV (see Appendix 1). The total dose will be calculated based on the patient's weight on Day 1 of each cycle (or up to 3 days before) with no upper limit.

If the timing of trastuzumab emtansine coincides with a holiday that precludes the procedure, the procedure should be performed within 3 business days of the scheduled date and, when possible, on the earliest following date, with subsequent protocol-specified procedures rescheduled accordingly.

The first infusion of trastuzumab emtansine will be administered over 90 minutes (±10 minutes). Infusions may be slowed or interrupted for patients experiencing infusion-associated symptoms. Vital signs must be assessed before and after dose administration. Following the initial dose, patients will be observed for at least 90 minutes for fever, chills, or other infusion-associated symptoms. If prior infusions were well tolerated (without any signs or symptoms of infusion reactions), subsequent doses of trastuzumab emtansine may be administered over 30 minutes (±10 minutes), with a minimum 30-minute observation period following infusion. Local health authority guidelines must be followed with regard to further observation and monitoring, if applicable.

Pre-medication for nausea and infusion reactions (e.g., acetaminophen or other analgesics, antihistamines such as diphenhydramine, or corticosteroids) may be given at the investigator's discretion.

# Capecitabine

Capecitabine will be administered twice a day, orally for 14 days followed by a 7-day rest period at the Dose Levels described in Section 3.1.1. Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Capecitabine doses can be delayed for up to 4 hours, while keeping the minimal interval of 8 hours between the doses.

Rounding of the dose, based on 150 and 500 mg strength tablets, will be allowed to the nearest dose per patient body surface area (BSA).

If a dose is missed, the patient should skip that dose. The patient should not double the dose during the next administration.

Guidelines for dosage modification and treatment interruption or discontinuation are provided in Section 5.1.

#### 4.3.2.2 For Patients with LA/mGC

#### Trastuzumab Emtansine

Trastuzumab emtansine will be administered on Day 1 qw at a dose of 2.4 mg/kg IV (see Appendix 1). The total dose will be calculated based on the patient's weight on Day 1 of each cycle (or up to 3 days before) with no upper limit.

Administration time and observation period are described in Section 4.3.2.1 for trastuzumab emtansine.

Guidelines regarding timing delays and infusion times are the same as for patients with mBC, as is the accepted pre-medication.

## Capecitabine

Capecitabine will be administered at a starting dose of 700 mg/m² bid, orally, for 14 days followed by a 7-day rest period (the dose level determined as the MTD in cohort 1, with de-escalation as described in section 3.1.1.3. Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Capecitabine doses can be delayed for up to 4 hours, while keeping the minimal interval of 8 hours between the doses.

If a dose is missed, the patient should skip that dose. The patient should not double the dose at the next administration.

Guidelines for dosage modification and treatment interruption or discontinuation are provided in Section 5.1.

# 4.3.3 INVESTIGATIONAL MEDICINAL PRODUCT ACCOUNTABILITY

All investigational medicinal products (IMPs) required for completion of this study (trastuzumab emtansine and capecitabine) will be provided by the Sponsor. The investigational site will acknowledge receipt of IMPs, using the interactive voice/web recognition system (IxRS) to confirm the shipment condition and content. Any damaged shipments will be replaced.

IMPs will be either disposed of at the study site according to the study site's institutional standard operating procedure or returned to the Sponsor with the appropriate documentation. The site's method of IMP destruction must be agreed upon by the Sponsor. The site must obtain written authorization from the Sponsor before any IMP is destroyed, and IMP destruction must be documented on the appropriate form.

Accurate records of all IMPs received at, dispensed from, returned to, and disposed of by the study site should be recorded on the Drug Inventory Log.

#### 4.3.4 Post-trial Access to Extension Study

Post-trial access to trastuzumab emtansine and capecitabine will be performed as described in Section 3.1.1, *Duration of Treatment and Patient Follow-Up*. If a patient decides to withdraw from the study, no post-trial access will be granted. Currently, the Sponsor does not have any plans to provide

other study interventions to patients after conclusion of the study or any earlier patient withdrawal.

# 4.4 CONCOMITANT AND EXCLUDED THERAPIES

## 4.4.1 PERMITTED THERAPY

Concomitant therapy and pre-medication are defined as non-IMPs.

Concomitant therapy includes any prescription medication, over-the-counter preparation, or herbal therapy between the 14 days preceding first treatment and the Study Treatment Discontinuation Visit. Afterwards, only anti-cancer therapies will be collected as part of the survival follow-up.

Pre-medication is allowed according to standard practice guidelines.

No pre-medication for the first infusion of trastuzumab emtansine is required; however, pre-medication is allowed at the investigator's discretion.

Concomitant use of erythropoiesis-stimulating agents is allowed if clinically indicated in accordance with local prescribing guidelines.

Palliative radiotherapy is permitted to treat pre-existing painful bone metastases or to treat brain metastases (for patients who have disease control outside of the brain). Please contact the Medical Monitor for approval. If the Medical Monitor cannot be reached because of time zone differences, radiotherapy may be administered, but the Medical Monitor should still be informed.

Other medications considered necessary for the patient's safety and wellbeing may be given at the discretion of the investigator. Use of bisphosphonates or denosumab is permitted for the control of bone pain, prevention and/or treatment of bony metastases, and treatment of osteoporosis. If bisphosphonates are required for the treatment of symptomatic malignancy-associated hypercalcemia, tumor assessments should be performed to assess for potential PD.

#### 4.4.2 PROHIBITED THERAPY

During the study, use of the therapies described below is prohibited until discontinuation of study treatment (collectively, these will be referred to as non-protocol therapy).

Any therapies intended for the treatment of cancer, other than trastuzumab emtansine, whether they are approved by national health authorities or experimental, including cytotoxic chemotherapy, immunotherapy, hormonal therapy (other than megestrol acetate), and biologic or targeted agents (other than granulocyte colony-stimulating factor and erythropoiesis-stimulating agents), are prohibited.

Radiotherapy for unequivocal PD is not permitted while on study treatment, with the exception of new brain metastases or isolated progression of previously treated brain lesions. Patients who have disease control outside of

the brain, defined as continued PR or CR of any duration, or SD for  $\geq 3$  months, but who have developed brain metastases that are treatable with radiation will be allowed to continue to receive study therapy until they either experience systemic progression of their disease and/or further progression in the brain that cannot be treated with additional radiation. Patients must not miss more than one cycle of study treatment for the treatment of their brain metastases and must have an ECOG performance status of 0, 1, or 2 to continue on therapy. The Medical Monitor should be informed before a decision is made to resume study treatment after radiotherapy for brain metastases.

# 4.5 STUDY ASSESSMENTS

All patients will be closely monitored for safety and tolerability during all cycles of therapy and at the safety follow-up visit:

- Visits will be based on a q3w cycle for mBC
- Visits will be based on a qw cycle for mGC

Study assessments are outlined in this section and in Appendix 1.

## 4.5.1 DESCRIPTION OF STUDY ASSESSMENTS

All patients will be closely monitored for safety and tolerability during all cycles of therapy and at the Study Treatment Discontinuation Visit. Patients should be assessed for toxicity prior to each dose; dosing will occur only if the clinical assessment and local laboratory test values are acceptable. Trastuzumab emtansine will be administered either in q3w cycles (patients with mBC) or qw cycles (patients with mGC) if no additional time is required for resolution of toxicity. Dose delays and dose reductions will be allowed for trastuzumab emtansine as outlined in Section 5.1.5.

If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend that precludes the procedure within the allotted window, the procedure should be performed on the nearest following date (i.e., within 3 business days).

# 4.5.1.1 Medical History and Demographic Data

Medical history includes clinically significant diseases, surgeries, cancer history (including prior cancer therapies and procedures), smoking history, use of alcohol and drugs of abuse, and all medications (e.g., prescription drugs, over-the-counter drugs, herbal/homeopathic remedies, nutritional supplements) used by the patient within 14 days prior to the screening visit.

Demographic data will include age, sex, and self-reported race/ethnicity (unless not allowed per local regulations).

# 4.5.1.2 Vital Signs

Vital signs will include measurements of weight, respiratory rate, heart rate, blood pressure, and temperature. Abnormal or significant changes to vital signs from baseline should be recorded as AEs, if appropriate.

# 4.5.1.3 Physical Examinations

A complete physical examination should include the evaluation of head, eye, ear, nose, and throat; cardiovascular; dermatological; musculoskeletal; respiratory; gastrointestinal; and neurological systems. Changes from baseline abnormalities should be recorded at each subsequent physical examination. New or worsened abnormalities should be recorded as AEs if appropriate.

As part of the tumor assessment, physical examinations should also include the evaluation of the presence and degree of enlarged lymph nodes, hepatomegaly, and splenomegaly.

Limited physical examinations will be symptom-directed.

# 4.5.1.4 Tumor and Response Evaluations

Measurable and unmeasurable disease must be documented at screening and re-assessed at each subsequent tumor evaluation. Tumor assessments with computed tomography (CT) or magnetic resonance imaging (MRI) scans of the chest, abdomen, and pelvis are to be performed as described in Appendix 1, Schedule of Assessment. CT or MRI of the brain and baseline radioisotope bone scan must be obtained at screening. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to first treatment the bone scan does not need to be repeated and non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Tumor assessments should include an evaluation of all known and/or suspected sites of disease, whenever possible. Patients should have lesions selected that can be evaluated at every tumor assessment. The same radiographic procedure used at screening must be used throughout the study (e.g., the same contrast protocol for CT scans). Response assessments will be assessed by the investigator, based on physical examinations, CT or MRI scans, and bone scans using RECIST v. 1.1 (see Appendix 3). In the event a positron emission tomography (PET)/CT scanner is used for tumor assessments, the CT portion of the PET/CT must meet criteria for diagnostic quality. For patients who continue study treatment after isolated brain progression, the frequency of follow-up scans is at the discretion of the investigator.

At the investigator's discretion, CT scans, MRI scans, and/or bone scans may be obtained at any time when clinically indicated or if PD is suspected. If a bone scan cannot be performed during the course of the study because of the unavailability of the Tc-99m isotope, the investigator may choose an alternative imaging modality (see Appendix 4).

Radiographic imaging should always be performed rather than clinical examination unless the lesion(s) being followed cannot be imaged but is assessable by clinical examination. In applying RECIST, documentation by color photography including a ruler to estimate the size of the lesion is recommended.

## 4.5.1.5 Laboratory Assessments

#### For Patients with mBC:

## **Local Laboratory Assessments:**

- Hematology, biochemistry, coagulation, urinalysis, and pregnancy testing
- Prospective or retrospective HER2 status. Patients will be enrolled based on local results.

## **Central Laboratory Assessments:**

- Retrospective HER2 status. Retrospective central confirmation will not impact the treatment decisions or primary endpoint of Phase I, Cohort 1 and will be used to validate efficacy analyses in Phase I and to define subgroups for efficacy analyses in the Randomized Phase II part of the study
- PK assays:
- Serum trastuzumab emtansine concentration and total trastuzumab using a validated immunoassay
- Serum capecitabine and 5-FU PK samples
- Plasma concentration of DM1 using a validated liquid chromatography electrospray tandem mass spectrometry (LC-MS/MS) method

## For Patients with mGC:

## **Local Laboratory Assessments:**

Hematology, biochemistry, coagulation, urinalysis, and pregnancy testing

#### **Central Laboratory Assessments:**

- Prospective HER2 status. Patients will be enrolled based on the central testing results
- PK assays:
- Serum trastuzumab emtansine concentration and total trastuzumab using a validated immunoassay
- Serum capecitabine and 5-FU PK samples
- Plasma concentration of DM1 using a validated LC-MS/MS method

# 4.5.1.6 Electrocardiograms

A 12-lead ECG should be obtained at baseline and be printed and kept with the patient's record.

#### 4.5.1.7 ECOG Performance Status

Performance status will be measured using the ECOG performance status scale (see Appendix 6).

It is recommended, where possible, that a patient's performance status be assessed by the same person throughout the study.

Performance status will be assessed according to the schedule of assessments (see Appendix 1).

## 4.5.1.8 ECHO/MUGA

ECHO is the preferred modality because of the global technetium (Tc-99m) shortage (see Appendix 4). The same method used at screening should be used throughout the study.

## 4.5.2 TIMING OF STUDY ASSESSMENTS

## 4.5.2.1 Screening and Pretreatment Assessments

Written informed consent for participation in the study must be obtained before performing any study-specific screening tests or evaluations. Informed Consent Forms for enrolled patients and for patients who are not subsequently enrolled will be maintained at the study site.

Once the patient has signed the Informed Consent Form, the investigator (or his or her designee) will call the IxRS to obtain the screening number for the patient prior to Cycle 1, Day 1.

Results of standard of care tests or examinations performed prior to obtaining informed consent and within 28 days prior to study start may be used; such tests do not need to be repeated for screening. Patients must have stable LFTs before the first dose of study drug.

All screening evaluations must be completed and reviewed to confirm that patients meet all eligibility criteria before study start. The investigator will maintain a screening log to record details of all patients screened and to confirm eligibility or record reasons for screening failure, as applicable.

Patients in Cohort 1 will not contribute to Phase II; however, they will be followed up until EOS. In the Randomized Phase II part, patients will be randomized in a 1:1 ratio to receive trastuzumab emtansine alone or the combination of trastuzumab emtansine and capecitabine prior to receiving the first dose of study medication.

The IxRS will be available 24 hours a day, 7 days a week. Detailed instructions regarding the IxRS will be provided to each study center. The screening numbers are to be allocated according to the specification document agreed with the IxRS provider.

Please see Appendix 1 for the schedule of screening assessments.

# 4.5.2.2 Assessments during Treatment

#### For Patients with mBC

Scheduled study visits are based on a q3w cycle, with Cycle 1 beginning at Day 1. All visits must occur within ± 3 business days from the scheduled date, unless otherwise noted in the schedule of assessments. All assessments will be performed on the day of the specified visit unless a time window is specified. Assessments scheduled on the day of study treatment administration should be performed prior to study treatment administration unless otherwise noted. If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend, it should be performed on the nearest following date (i.e., within 3 business days).

Local laboratory assessments scheduled for Day 1 of all cycles must be performed within 72 hours prior to study treatment administration unless otherwise specified. Results of local laboratory assessments must be reviewed and the review documented prior to study treatment administration.

Please see Appendix 1 for the schedule of treatment period assessments.

#### For Patients with mGC

Scheduled study visits are based on a qw cycle, with Cycle 1 beginning at Day 1. All visits must occur within ± 3 business days from the scheduled date, unless otherwise noted in the schedule of assessments. All assessments will be performed on the day of the specified visit unless a time window is specified. Assessments scheduled on the day of study treatment administration should be performed prior to study treatment administration unless otherwise noted. If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend, it should be performed on the nearest following date (i.e., within 3 business days).

Local laboratory assessments scheduled for Day 1 of all cycles must be performed within 72 hours prior to study treatment administration unless otherwise specified. Results of local laboratory assessments must be reviewed and the review documented prior to study treatment administration.

Please see Appendix 1 for the schedule of treatment period assessments.

## 4.5.2.3 Assessments at Study Completion/Early Termination Visit

Patients may remain on study treatment until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor. Patients who discontinue study treatment will be followed up until EOS and will be asked to return to the clinic approximately 28–42 days after the last study treatment administration for the safety follow-up visit.

Please see Appendix 1 for assessments to be performed at the safety followup visit.

73

# 4.5.2.4 Follow-up Assessments

After the Study Treatment Discontinuation Visit, all patients (regardless of reason for discontinuation) will have survival status and anti-cancer therapies recorded and will be followed for all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or dies, or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration.

Patients who discontinue study drugs for any reason other than PD or withdrawal of consent (e.g., an AE) will continue to be followed according to the tumor assessment schedule until withdrawal of consent, death, or EOS, whichever occurs first.

After the study treatment completion/early termination visit, AEs should be followed as outlined in Section 5.5 and 5.6.

Please see Appendix 1 for the schedule of follow-up assessments.

# 4.5.2.5 Assessments at Unplanned Visits

In case unplanned visits are required, electronic Case Report Form (eCRF) pages will be available to report the information collected during those visits.

# 4.6 PATIENT AND STUDY DISCONTINUATION

# 4.6.1 PATIENT DISCONTINUATION

Patients have the right to withdraw from the study at any time for any reason. The investigator has the right to discontinue a patient from study treatment or from the study for any medical condition that the investigator determines may jeopardize the patient's safety if he or she continues in the study, for reasons of non-compliance (e.g., missed doses, visits), if the patient becomes pregnant, or if the investigator determines it is in the best interest of the patient.

Patients must be withdrawn from study treatment if they become pregnant or experience PD defined using RECIST v. 1.1 (<u>Appendix 3</u>). The exception to this is patients who develop isolated progression in the brain as described in <u>Appendix 3</u>.

Details of discontinuation due to toxicity are given in Section 5.1.

Patients who discontinue from study treatment prematurely for any of the above reasons will continue to be followed according to Section 4.5.2.4 "Follow-Up Assessments". The primary reason for discontinuation must be recorded on the appropriate eCRF page.

#### 4.6.2 STUDY DISCONTINUATION

Sections 3.1.1 and 3.2 describe the EOS definition and discontinuation of study treatment. Prior to that, the Sponsor has the right to terminate this study **Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd**Protocol MO28230, Version 3, 30 June 2014

at any time. Reasons for terminating the study may include, but are not limited to, the following:

- The incidence or severity of AEs in this or other studies indicates a potential health hazard to patients
- Patient enrollment is unsatisfactory
- Data recording is inaccurate or incomplete.

# 5. ASSESSMENT OF SAFETY

Overall safety will be assessed on an ongoing basis during the conduct of the study.

# 5.1 SAFETY PLAN

The safety plan for patients receiving trastuzumab emtansine is based on the toxicities of trastuzumab emtansine observed in nonclinical studies; the toxicities related to its components (trastuzumab and maytansine, the parent drug of DM1) observed in clinical studies; and the clinical experience with this molecule in completed and ongoing studies. Please refer to the trastuzumab emtansine and capecitabine (Xeloda®) Investigator's Brochures for the most recent information.

All patients will be monitored closely for toxicity. The important safety issues anticipated in this trial, as well as measures intended to avoid or minimize such toxicities, are outlined in the following sections.

## 5.1.1 RISKS ASSOCIATED WITH TRASTUZUMAB EMTANSINE

Full details regarding the clinical safety of trastuzumab emtansine are presented in Sections 5 and 6 of the Investigator's Brochure.

# 5.1.1.1 Cardiotoxicity

Patients treated with trastuzumab emtansine are at increased risk of developing left ventricular dysfunction. LVEF < 40% has been observed in patients treated with trastuzumab emtansine. Patients without significant cardiac history and with an LVEF  $\ge$  50% determined by ECHO or MUGA scan are eligible for study participation. LVEF will be monitored at screening and regularly throughout the study until the assessment at the safety follow-up visit. Patients with symptomatic cardiac dysfunction will be discontinued from study treatment. Asymptomatic LVEF declines will be handled according to the algorithm shown in Figure 6. Treatment with trastuzumab emtansine has not been studied in patients with LVEF < 50%.

# 5.1.1.2 Hematologic Toxicity (Thrombocytopenia)

Thrombocytopenia, or decreased platelet counts, was reported in patients in clinical trials of trastuzumab emtansine. The majority of these patients had Grade 1 or 2 events ( $\geq 50,000/\text{mm}^3$ ), with the nadir occurring by Day 8 and generally improving to Grade 0 or 1 ( $\geq 75,000/\text{mm}^3$ ) by the next scheduled

dose. In clinical trials, the incidence and severity of thrombocytopenia were higher in Asian patients. Severe cases of both non-fatal and fatal hemorrhagic events including central nervous system hemorrhage have been reported in clinical trials with trastuzumab emtansine; these events were independent of the patients' ethnicity. In some of the observed cases the patients were also receiving anti-coagulation therapy. The need for platelet transfusions has been reported.

Patients with thrombocytopenia and on anti-coagulant treatment have to be monitored closely during treatment with trastuzumab emtansine. Platelet counts will be monitored prior to each trastuzumab emtansine dose.

Use of erythropoiesis-stimulating agents will be allowed as consistent with prescribing guidelines. Transfusion of red blood cells and/or platelets will be allowed according to and at the discretion of the treating physician.

# 5.1.1.3 Hepatotoxicity

Hepatotoxicity, predominantly in the form of asymptomatic increases in the concentrations of serum transaminases (Grade 1–4 transaminitis), has been observed in patients while on treatment with trastuzumab emtansine in clinical trials. Transaminase elevations were generally transient. A cumulative effect of trastuzumab emtansine on transaminases has been observed; elevated transaminases improved to Grade 1 or normal within 30 days of the last dose of trastuzumab emtansine in the majority of the patients. Serious hepatobiliary disorders, including nodular regenerative hyperplasia (NRH) of the liver and some resulting in fatal liver failure, have been observed in patients treated with trastuzumab emtansine in clinical trials. Some of the observed cases may have been confounded by comorbidities and/or concomitant medications with known hepatotoxic potential. Liver function should be monitored before initiation of treatment and each trastuzumab emtansine dose.

Trastuzumab emtansine has not been studied in patients with serum transaminases  $> 2.5 \times \text{ULN}$  or total bilirubin  $> 1.5 \times \text{ULN}$  before initiation of treatment. Trastuzumab emtansine treatment in patients with serum transaminases  $> 3 \times \text{ULN}$  and concomitant total bilirubin  $> 2 \times \text{ULN}$  should be permanently discontinued.

Cases of NRH of the liver have been identified from liver biopsies in patients presenting with signs and symptoms of portal hypertension. NRH was also observed in one fatal case of hepatic failure. NRH is a rare liver condition characterized by widespread benign transformation of hepatic parenchyma into small regenerative nodules; NRH may lead to non-cirrhotic portal hypertension. Diagnosis of NRH can only be confirmed by histopathology. NRH should be considered in patients who develop clinical symptoms of portal hypertension and/or a cirrhosis-like pattern seen on CT scan of the liver but with normal transaminases and no other manifestations of cirrhosis or liver failure following long-term treatment with trastuzumab emtansine. Upon diagnosis of NRH, trastuzumab emtansine treatment must be permanently discontinued.

# 5.1.1.4 Pulmonary Toxicity

Cases of interstitial lung disease (ILD), including pneumonitis, some leading to acute respiratory distress syndrome or fatal outcome, have been reported in clinical trials with trastuzumab emtansine. Signs and symptoms include dyspnea, cough, fatigue, and pulmonary infiltrates. These events may or may not occur as sequelae of infusion reactions. Treatment has included administration of steroids and oxygen, and study drug discontinuation. Patients with dyspnea at rest due to complications of advanced malignancy and comorbidities may be at increased risk of pulmonary events.

Treatment with trastuzumab emtansine has to be permanently discontinued in patients who are diagnosed with ILD or pneumonitis.

## 5.1.1.5 Infusion-related Reactions/Hypersensitivity

Infusion-related reactions characterized by one or more of the following symptoms, flushing, chills, pyrexia, dyspnea, hypotension, wheezing, bronchospasm, and tachycardia may occur with the administration of monoclonal antibodies and have been reported with trastuzumab emtansine. In general, these symptoms were not severe. In most patients, these reactions resolved over the course of several hours to a day after the infusion was terminated. Patients should be observed closely for infusion-related reactions, especially during the first infusion.

Patients should be observed closely for hypersensitivity. Serious, allergic/anaphylactic-like reactions have been observed in clinical trials with treatment of trastuzumab emtansine. Administration of trastuzumab emtansine will be performed in a setting with access to emergency facilities and staff who are trained to monitor and respond to medical emergencies. Patients will be observed closely for infusion-related/hypersensitivity during and after each trastuzumab emtansine infusion for a minimum of 90 minutes after the first infusion and for a minimum of 30 minutes after subsequent infusions in the absence of infusion-related AEs. Pre-medication is allowed according to standard practice guidelines. In the event of a true hypersensitivity reaction (in which severity of reaction increases with subsequent infusions), trastuzumab emtansine treatment must be permanently discontinued. Patients who experience a Grade  $\geq$  3 allergic reaction or acute respiratory distress syndrome will be discontinued from study treatment.

# 5.1.1.6 Neurotoxicity

DM1, an anti-microtubule agent, can potentially cause peripheral neuropathy. Peripheral neuropathy, mainly Grade 1 and predominantly sensory, has been reported in clinical trials of trastuzumab emtansine. Treatment with trastuzumab emtansine should be temporarily discontinued in patients experiencing Grade 3 or 4 peripheral neuropathy until symptoms resolve or improve to  $\leq$  Grade 2. Patients should be examined for signs of peripheral neuropathy prior to each dose of trastuzumab emtansine. Patients who experience Grade  $\geq$  3 neurotoxicity in the form of peripheral neuropathy that

does not resolve to Grade ≤ 2 within 42 days after last dose received will be discontinued from study treatment.

#### 5.1.1.7 Extravasation

In trastuzumab emtansine clinical studies, reactions secondary to extravasation have been observed. These reactions were usually mild and comprised erythema, tenderness, skin irritation, pain, or swelling at the infusion site. Rare reports of more severe events such as cellulitis, pain (tenderness and burning sensation), and skin irritation have been received as part of the continuing surveillance of trastuzumab emtansine safety. These reactions have been observed more frequently within 24 hours of infusion. Specific treatment for trastuzumab emtansine extravasation is unknown at this time. The infusion site should be closely monitored for possible subcutaneous infiltration during drug administration.

### 5.1.1.8 Trastuzumab Emtansine Dose Modification

Trastuzumab emtansine dose modifications are described in Section 5.1.5.1.

#### 5.1.2 RISKS ASSOCIATED WITH CAPECITABINE

Patients treated with capecitabine should be carefully monitored for toxicity. Most AEs are reversible and do not require permanent discontinuation of therapy (please refer to the Xeloda® SmPC for more information).

The spectrum of cardiotoxicity observed with capecitabine is similar to that of other fluorinated pyrimidines. This includes myocardial infarction, angina, dysrhythmias, cardiac arrest, cardiac failure and electrocardiographic changes. These AEs may be more common in patients with a prior history of coronary artery disease.

A rare, unexpected, severe toxicity (e.g. stomatitis, diarrhea, neutropenia, and neurotoxicity) associated with 5-FU has been attributed to deficiency of DPD activity. Therefore, a link between decreased levels of DPD and increased, potentially fatal, toxic effects of 5-FU cannot be excluded.

Capecitabine can induce hand-foot syndrome (palmar-plantar erythrodysesthesia or chemotherapy-induced acral erythema), which is a cutaneous toxicity. For patients receiving capecitabine monotherapy in the metastatic setting, the median time to onset was 79 days (range 11–360 days), with a severity range of Grades 1 to 3. Grade 1 hand-foot syndrome is defined by numbness, dysesthesia/paresthesia, tingling or erythema of the hands and/or feet and/or discomfort which does not disrupt normal activities. Grade 2 is defined as painful erythema and swelling of the hands and/or feet and/or discomfort affecting the patient's activities of daily living (ADL). Grade 3 is defined as moist desquamation, ulceration, blistering or severe pain of the hands and/or feet and/or severe discomfort that causes the patient to be unable to work or perform ADL. If Grade 2 or 3 hand-foot syndrome occurs, administration of capecitabine should be interrupted until the event resolves or decreases in intensity to Grade 1. Following Grade 3 hand-foot syndrome, subsequent doses of capecitabine should be decreased.

Capecitabine can induce hyperbilirubinemia. Administration of capecitabine should be interrupted if treatment-related elevations in bilirubin of > 3.0 × ULN or treatment-related elevations in hepatic aminotransferases (ALT/AST) of Grade ≥ 2 occur.

Capecitabine can induce severe skin reactions such as Stevens-Johnson syndrome and toxic epidermal necrolysis. Capecitbaine should be permanently discontinued in patients who experience a severe skin reaction during treatment.

# 5.1.3 RISKS ASSOCIATED WITH TRASTUZUMAB EMTANSINE AND CAPECITABINE COMBINATION

The two DLTs observed in Phase I, Cohort 1 (in mBC) were grade 3 vomiting in one patient and grade 3 elevated AST and ALT in one patient (see Section 3.1.1.2). Both patients were treated at dose level 1 (capecitabine 750 mg/m² bid, days 1–14) in combination with trastuzumab emtansine 3.6 mg/kg q3w). During Phase I in LA/mGC, DLTs for the combination of trastuzumab emtansine and capecitabine will be observed during Cycle 1 (Days 1–21) of this study. The combination treatment must be considered as a new treatment during Cycle 1, and no individual dose reduction will be allowed during Cycle 1; the general DLT rules will be used instead. Interruptions can be made due to toxicities considered by the investigator to be related to capecitabine. Grade 2–4 toxicities should be interrupted until resolved to Grade 0–1. For Grade 4 toxicities, consideration to discontinue treatment with capecitabine will be made with the adjudication of the SC.

# 5.1.4 DEFINITION OF DOSE-LIMITING TOXICITY

DLTs will be observed during Cycle 1 (Day 1–21). Please refer to the Xeloda<sup>®</sup> SmPC for recommendations on dose reduction in subsequent cycles.

# **Definition of DLT:**

#### <u>Hematologic</u>

- 1. Uncomplicated Grade 4 thrombocytopenia that does not recover to ≥ 75,000/MI before Day 21
- 2. Thrombocytopenia (any grade) complicated with clinically significant bleeding requiring medical intervention, such as platelet transfusion or cauterization. However, patients with Grade 1 or 2 epistaxis may have cauterization and this should not be considered as a DLT.
- 3. Grade 4 neutropenia lasting > 7 consecutive days
- 4. Febrile neutropenia with an ANC of < 1,000 cells/mm<sup>3</sup>

## Non-hematologic

- 5. Grade ≥ 3 diarrhea that does not decrease to Grade ≤ 2 after 24 hours of starting recommended anti-diarrheal treatment
- 6. Grade 3 hand-foot syndrome (Grade 4 not applicable)

7. Any other treatment-related toxicity Grade ≥ 3 prohibiting the start of the second cycle on Day 22 (3 weeks cycle length plus 1 day)

NOTE: If a Grade 2 event requires a dose delay, it will not be considered as a DLT. However, if the toxicity does not resolve to Grade 1 or baseline by Day 42, this requires discontinuation and will be considered as a DLT.

8. Grade 2 toxicity requiring interruption of treatment for > 14 days

NOTE: Patients experiencing Grade ≥ 3 hand-foot syndrome, diarrhea, mucositis, or febrile neutropenia with ANC < 500 cells/mm<sup>3</sup> during Cycle 1 must be tested for DPD deficiency (a central laboratory will be appointed). The SC will adjudicate in cases of DLTs that are not covered by the existing DLT criteria.

- 9. Having taken < 14 full doses of capecitabine due to toxicity
- Patient not able to receive 100% of the dose level going into Cycle 2, Day 1

## 5.1.5 MANAGEMENT OF SPECIFIC ADVERSE EVENTS

### 5.1.5.1 Trastuzumab Emtansine Dose Modification

Patients should be assessed for toxicity prior to each dose; dosing will occur only if the clinical assessment and laboratory test values are acceptable.

Dose delays and reductions are designed to maximize treatment for those who derive clinical benefit from treatment while ensuring patient safety. Dose delays for trastuzumab emtansine-related toxicity other than those specified below (i.e., infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, cardiotoxicity, and ILD or pneumonitis) are as follows:

- If significant trastuzumab emtansine-related toxicities (other than infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, and cardiotoxicity) have not recovered to Grade 1 or baseline, the next scheduled dose may be delayed for up to 42 days from the last dose received. "Significant" and "related" will be based on the judgment of the investigator (in consultation with the Sponsor's Medical Monitor or designee when appropriate). For example, alopecia even if considered related would most likely not be considered to be significant. Fatigue may or may not be considered either related or significant.
- In general, when the significant and related toxicity (or any other toxicity that the investigator chooses to delay dosing for) resolves to Grade 1 or baseline, the patient may resume trastuzumab emtansine if the delay has not exceeded 42 days from the last received dose. Patients should be reevaluated qw during the delay, whenever possible. If dosing resumes, the patient may receive trastuzumab emtansine either at the same dose level as before or at one dose level lower (see Table 2 and Table 3), at the discretion of the investigator. Subsequent cycles should remain the same (q3w or qw), and patients should be assessed for toxicity.

- If a patient requires a dose reduction, dosing will be reduced by one dose level, per Table 2or Table 3. No dose re-escalation will be allowed.
- If toxicity does not resolve within 42 days from the last dose received, the patient will be discontinued from study treatment and will be followed for PD and survival outcome as described in Section 5.5.
- Patients who experience a Grade 3 or 4 hematologic event should be checked at least weekly for recovery. If values do not recover to baseline or Grade ≤ 1 within 42 days from the last dose received, the patient will be discontinued from study treatment.

Table 2 Dose Reduction for Trastuzumab Emtansine (Patients with mBC)

| Dose Level | q3w Schedule |
|---------------------------------------------|---------------------|
| Dose Level | ' |
| 0 | 3.6 mg/kg |
| - 1 | 3.0 mg/kg |
| - 2 | 2.4 mg/kg |
| Indication for<br>further dose<br>reduction | Off study treatment |

q3w = every 3 weeks

Table 3 Dose Reductions for Trastuzumab Emtansine (Patients with mGC)

| | qw Schedule |
|---------------------------------------|-------------|
| Dose Level | |
| 0 | 2.4 mg/kg |
| - 1 | 2.0 mg/kg |
| - 2 | Off study |
| Indication for further dose reduction | Off study |

qw = weekly

In case of toxicities requiring the discontinuation of trastuzumab emtansine, the patient will be followed-up until the EOS.

Protocol requirements for specific toxicities are outlined below.

# 5.1.5.1.1 Trastuzumab Emtansine Dose Modification for Thrombocytopenia

Platelet counts should be obtained no less frequently than weekly to evaluate recovery whenever any of the events listed below occurs. If platelet counts do not recover to Grade ≤ 1 within 42 days from the last dose received, the patient will be discontinued from study treatment.
No re-escalation of the trastuzumab emtansine dose is allowed.

Note: although complete blood counts with platelets are required within 72 hours prior to study treatment administration at each cycle, the investigator may monitor platelet counts (or any other laboratory test) more frequently as clinically indicated.

In the event of decreased platelet count to Grade 3 ( $< 50,000/\text{mm}^3$ ), do not administer trastuzumab emtansine until platelet counts recover to Grade 1 ( $\ge 75,000/\text{mm}^3$ ), then treat at the same dose level.

Patients receiving trastuzumab emtansine who experience a first Grade 4 thrombocytopenia event may, after adequate recovery to a platelet count of Grade ≤ 1 or baseline, continue treatment with trastuzumab emtansine at a dose of 3 mg/kg in subsequent treatment cycles. Patients at the 3 mg/kg dose level who experience a Grade 4 thrombocytopenia event may, after adequate recovery as defined above, continue treatment with trastuzumab emtansine at a dose of 2.4 mg/kg in subsequent treatment cycles. Patients who experience a Grade 4 thrombocytopenia event at the 2.4 mg/kg dose level will be discontinued from study treatment. A dose delay of up to 42 days from the patient's last dose received is permitted.

### 5.1.5.1.2 Trastuzumab Emtansine Dose Modification for Hepatotoxicity

### 5.1.5.1.2.1 Concurrent elevations of ALT/AST and bilirubin meeting Hy's Law laboratory criteria

Regardless of dose level, trastuzumab emtansine must be <u>permanently</u> <u>discontinued</u> in patients with ALT and/or AST > 3 × ULN and concurrent increase of total bilirubin to > 2 × ULN. All relevant hepatic laboratory tests performed (including AST, ALT, total bilirubin, alkaline phosphatase, activated partial thromboplastin time [aPTT], INR, and albumin) will be entered into the clinical database.

#### 5.1.5.1.2.2 Nodular regenerative hyperplasia

Trastuzumab emtansine must be permanently discontinued in patients who are diagnosed with NRH.

### 5.1.5.1.2.3 Transaminase elevations or bilirubin elevation requiring dose adjustment

Patients who experience a Grade 3 elevation of liver function should be checked twice weekly for the recovery of transaminases and/or total bilirubin. If a patient's transaminases and/or total bilirubin do not recover according to Table 4 and Table 5, within 42 days from the patient's last dose received, the patient will be discontinued from study treatment.

No re-escalation of the trastuzumab emtansine dose is allowed.

Table 4 and Table 5 describe the dose modification guidelines for increases in serum bilirubin and transaminases, respectively.

Table 4 Trastuzumab Emtansine Dose Modification: Total Serum Bilirubin

| Grade 2 | Grade 3 | Grade 4 |
|---|---|---|
| (> 1.5 to ≤ 3 × ULN) | (> 3 to ≤ 10 × ULN) | (> 10 × ULN) |
| Do not administer trastuzumab emtansine until total bilirubin recovers to Grade ≤ 1, and then treat at the same dose level | Do not administer trastuzumab emtansine until total bilirubin recovers to Grade ≤ 1 and then reduce one dose level | Discontinue<br>trastuzumab<br>emtansine |

ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

Table 5 Trastuzumab Emtansine Dose Modification: Serum ALT or AST

| Grade 2 | Grade 3 | Grade 4 |
|---|---|---|
| (> 3 to ≤ 5 × ULN) | (> 5 to ≤ 20 × ULN) | (> 20 × ULN) |
| Treat at the same dose level | Do not administer trastuzumab<br>emtansine until AST/ALT<br>recovers to Grade ≤ 2, and<br>then reduce one dose level | Discontinue<br>trastuzumab<br>emtansine |

ALT = alanine transaminase; AST = aspartate transaminase; ULN = upper limit of normal. Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

#### **5.1.5.1.3** Trastuzumab Emtansine Dose Modification for Neurotoxicity

Patients receiving trastuzumab emtansine who experience Grade 3 or 4 peripheral neuropathy that does not resolve to Grade ≤ 2 within 42 days after the last dose received will be discontinued from study treatment.

### 5.1.5.1.4 Trastuzumab Emtansine Dose Modification for Cardiotoxicity

Patients without significant cardiac history and with a baseline LVEF  $\geq$  50% as determined by ECHO or MUGA scan are eligible for study participation. Ejection fractions will be monitored during the last week of Cycle 1, Cycle 3 and every third cycle thereafter until the assessment at the safety follow-up visit.

Figure 6 summarizes the management of trastuzumab emtansine on the basis of measured LVEF and changes in LVEF from baseline in patients. If the LVEF is reported as a range, the median of the range should be taken. If an investigator is concerned that an AE may be related to cardiac dysfunction, an additional LVEF measurement may be performed. Trastuzumab emtansine

will be discontinued in any patient who develops symptomatic CHF. CHF should be treated and monitored according to standard medical practice.

The decision to stop or continue trastuzumab emtansine should be based on the algorithm shown in Figure 6. Trastuzumab emtansine must be discontinued in all patients for whom a confirmed drop of LVEF to below 40% is documented (with a repeat assessment within 21 days). For patients whose LVEF drops to values between 40% and 45% with an absolute decrease in LVEF of  $\geq$  10% points from baseline, trastuzumab emtansine should be held. For these patients, the LVEF should be repeated in 21 days, and trastuzumab emtansine should be discontinued if the LVEF has not recovered to within 10% absolute difference below baseline. If clinically significant cardiac dysfunction or cardiac failure develops or persists or if significant medical management is required to maintain ejection fraction, the patient should be discontinued from study treatment.

Figure 6 Algorithm for Continuation and Discontinuation of Trastuzumab Emtansine Based on Left Ventricular Ejection Fraction Assessments in Patients



CHF = congestive heart failure; LVEF = left ventricular ejection fraction.

Note: LVEF assessment results must be reviewed before the next scheduled trastuzumab emtansine infusion.

- <sup>a</sup> LVEF can be repeated within 21 days, and trastuzumab emtansine should be discontinued if LVEF < 40% is confirmed. Trastuzumab emtansine should be held while the repeat LVEF is obtained.
- b After a second consecutive confirmatory result, trastuzumab emtansine should be discontinued if the LVEF is confirmed to be ≥ 10% points below baseline or if medical management was required to correct the LVEF.

## 5.1.5.1.5 Trastuzumab Emtansine Dose Modification/Management for Infusion-related Reactions, Hypersensitivity Reactions

Trastuzumab emtansine treatment should be interrupted in patients with severe infusion-related reactions. Trastuzumab emtansine treatment should be permanently discontinued in the event of life-threatening infusion-related reactions.

Infusion of trastuzumab emtansine should be interrupted for patients who develop dyspnea or clinically significant hypotension.

The infusion should be slowed to  $\leq 50\%$  or interrupted for patients who experience any other infusion-related symptoms. When the patient's symptoms have completely resolved, the infusion may be continued at  $\leq 50\%$  of the rate prior to the reaction and increased in 50% increments every 30 minutes as tolerated. Infusions may be restarted at the full rate during the next cycle.

Patients who experience trastuzumab emtansine infusion-related temperature elevations to > 38.5°C and/or other infusion-related symptoms may be treated symptomatically with acetaminophen and/or diphenhydramine hydrochloride. Serious infusion-related events manifested by dyspnea, hypotension, wheezing, bronchospasm, tachycardia, reduced oxygen saturation, or respiratory distress should be managed with supportive care, such as oxygen, beta agonists, antihistamines, antipyretics, or corticosteroids at the investigator's discretion. Pre-medication with corticosteroids, antihistamines, and antipyretics may be used before subsequent infusions of trastuzumab emtansine at the investigator's discretion. Patients should be monitored until complete resolution of symptoms. In the event of a true hypersensitivity reaction (i.e., if the severity of reaction increases with subsequent infusions), trastuzumab emtansine treatment must be permanently discontinued. Patients who experience a Grade ≥ 3 hypersensitivity reaction or acute respiratory distress syndrome (ARDS) will be discontinued from the study.

Patients who experience a severe delayed infusion reaction will be discontinued from study treatment.

### 5.1.5.1.6 Trastuzumab Emtansine Dose Modification for Pulmonary Toxicity

Cases of ILD, including pneumonitis (including severe, life-threatening cases) and some leading to ARDS or fatal outcome have been reported with trastuzumab emtansine. Treatment with trastuzumab emtansine has to be permanently discontinued in patients who are diagnosed with ILD or pneumonitis.

### 5.1.5.1.7 Trastuzumab Emtansine Dose Modification for Extravasation

During the clinical development of trastuzumab emtansine, reactions secondary to extravasation have been observed. These reactions were usually mild and consisted of erythema, tenderness, skin irritation, pain or swelling at the infusion site. Although trastuzumab emtansine is not considered as a vesicant, close monitoring of the infusion site for possible subcutaneous infiltration during drug administration is recommended.

#### 5.1.5.2 Capecitabine Dosage Modification

#### Phase I: Patients with mBC

The dose of capecitabine can be modified from Cycle 2 onwards if considered appropriate by the investigator (please refer to the Xeloda® SmPC for recommendations).

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued in patients with mBC.

During the Randomized Phase II part of the study, the dose of capecitabine will be modified according to the Xeloda® SmPC.

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued in patients with mBC.

#### Phase I: Patients with mGC

The dose of capecitabine can be modified from cycle 2 onwards if considered appropriate by the investigator (please refer to Xeloda® SmPC for recommendations).

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued (see Section 3.1.1).

#### 5.2 SAFETY PARAMETERS AND DEFINITIONS

Safety assessments will consist of monitoring and recording protocol-defined AEs and SAEs; measurement of protocol-specified hematology, clinical chemistry, and urinalysis variables; measurement of protocol-specified vital signs; and other protocol-specified tests that are deemed critical to the safety evaluation of the study drug(s).

The Sponsor or its designee is responsible for reporting relevant SAEs to the Competent Authority, other applicable regulatory authorities, and participating investigators, in accordance with International Conference on Harmonisation (ICH) guidelines, FDA regulations, European Clinical Trials Directive (Directive 2001/20/EC), and/or local regulatory requirements.

The Sponsor or its designee is responsible for reporting unexpected fatal or life-threatening events associated with the use of the study drug to the regulatory agencies and competent authorities by telephone or fax within 7 calendar days after being notified of the event. The Sponsor or its designee will report other relevant SAEs associated with the use of the study medication to the appropriate competent authorities (according to local guidelines), investigators, and central Institutional Review Boards/Ethics Committees (IRBs/ECs) by a written safety report within 15 calendar days of notification.

#### **ADVERSE EVENTS** 5.2.1

According to the ICH Guideline for Good Clinical Practice, an AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any of the following:

Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product

- Any new disease or exacerbation of an existing disease (a worsening in the character, frequency, or severity of a known condition), except as described in Section 5.3.5.7
- Recurrence of an intermittent medical condition (e.g., headache) not present at baseline
- Any deterioration in a laboratory value or other clinical test (e.g., ECG, X-ray) that is associated with symptoms or leads to a change in study treatment or concomitant treatment or discontinuation from study drug
- AEs that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment (e.g., screening invasive procedures such as biopsies)

## 5.2.2 SERIOUS ADVERSE EVENTS (IMMEDIATELY REPORTABLE TO THE SPONSOR)

A SAE is any AE that meets any of the following criteria:

- Fatal (i.e., the AE actually causes or leads to death)
- Life-threatening (i.e., the AE, in the view of the investigator, places the patient at immediate risk of death)

This does not include any AE that had it occurred in a more severe form or was allowed to continue might have caused death.

- Requires or prolongs inpatient hospitalization (see Section 5.3.5.8)
- Results in persistent or significant disability/incapacity (i.e., the AE results in substantial disruption of the patient's ability to conduct normal life functions)
- Congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug
- Significant medical event in the investigator's judgment (e.g., may jeopardize the patient or may require medical/surgical intervention to prevent one of the outcomes listed above)

The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an AE (rated as mild, moderate, or severe, or according to NCI CTCAE criteria; see Section 5.3.3); the event itself may be of relatively minor medical significance (such as severe headache without any further findings).

Severity and seriousness need to be independently assessed for each AE recorded on the eCRF.

SAEs are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2 for reporting instructions).

### 5.2.3 PROTOCOL-DEFINED EVENTS OF SPECIAL INTEREST/NON-SERIOUS EXPEDITED ADVERSE EVENTS

Non-serious AESIs are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event

(see Section 5.4.2 for reporting instructions) regardless of the attribution of causality. AESIs for this study include the following:

Potential drug-induced liver injury

Any case of potential drug-induced liver injury as assessed by laboratory criteria for Hy's law will be considered as a protocol-defined event of special interest and will need to be reported to the Sponsor expeditiously.

The following laboratory abnormalities define potential Hy's law cases:

AST and/or ALT elevations that are > 3 × ULN with concurrent elevation
of total bilirubin > 2 × ULN (or clinical jaundice if total bilirubin measures
are not available), except in patients with documented Gilbert's syndrome.
For patients with Gilbert's syndrome, elevation of direct bilirubin > 2 ×
ULN should be used instead

Suspected transmission of an infectious agent by the study drug:

 Defined as any organism, virus, or infectious particle (e.g., prion protein transmitting transmissible spongiform encephalopathy), both pathogenic and non-pathogenic. A transmission of an infectious agent may be suspected from clinical symptoms or laboratory findings indicating an infection in a patient exposed to a medicinal product. This term ONLY applies when a contamination of the study drug is suspected, NOT for infections supported by the mode of action, e.g., immunosuppression.

#### 5.2.4 Pregnancy and Contraception

ICH M3 guidance requires precautions to be taken to minimize risk to fetus or embryo when including women of childbearing potential in clinical studies. These precautions include the use of highly effective contraceptive measures, excluding pregnancy at baseline (serum test), continued pregnancy monitoring, and continued pregnancy testing for up to 7 months following last dose of study drug (follow-up period based on PK considerations).

Trastuzumab, a component of trastuzumab emtansine, can cause fetal harm when administered to a pregnant woman; postmarketing case reports indicate that its use during pregnancy increases the risk for oligohydramnios during the second and third trimester. Trastuzumab has also been associated with fetal pulmonary hypoplasia, skeletal abnormalities, and neonatal death (see the Herceptin® Package Insert). There are no clinical studies of trastuzumab in pregnant women. Immunoglobulin G (IgG) is known to cross the placental barrier.

Therefore, trastuzumab emtansine should be not used during pregnancy. Women of childbearing potential (who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy) and men with partners of childbearing potential must agree to use a highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the patient and/or partner.

Methods of birth control which result in a low failure rate (i.e., < 1% per year) when used consistently and correctly are considered highly effective forms of

contraception. The use of the following non-hormonal methods of contraception is acceptable:

- True abstinence, when this is the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, and symptothermal post ovulation methods) and withdrawal are not acceptable methods of contraception.
- Male sterilization (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female patients, the vasectomized male partner should be the sole partner.

Alternatively, use of two of the following effective forms of contraception is acceptable:

- Placement of intrauterine device (IUD) or intrauterine system (IUS).
   Consideration should be given to the type of device being used, as there are higher failure rates for certain types (e.g., steel or copper wire).
- Condom with spermicidal foam/gel/film/cream/suppository
- Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

The use of barrier contraceptives should always be supplemented with the use of a spermicide. The following should be noted:

- Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection.
- However, spermicides alone are ineffective at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

It should be noted that two forms of effective contraception are required. A double barrier method, defined as condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, is acceptable.

Contraception is not a requirement in the case of any of the following:

- The female patient or female partner of a male patient is considered not to be of childbearing potential: if she is postmenopausal, defined by amenorrhea of ≥ 12 months duration in a woman > 45 years old; or is ≥ 40 years of age and has had amenorrhea of ≥ 24 months duration; or has undergone surgical sterilization (hysterectomy and/or bilateral oophorectomy)
- The male patient or male partner of a female patient is surgically sterilized

For male patients with a female partner of childbearing potential, cooperation of female partner is required (i.e., use of two forms of contraception as stated above) during the study and for at least 7 months following the last dose of study treatment when a highly effective form of contraception is not appropriate.

Based on PK considerations, contraception must continue for the duration of study treatment and for at least 7 months after the last dose of study treatment.

A female patient or partner of a male patient who becomes pregnant during the study must be instructed to stop taking the study medication and immediately inform the investigator. The investigator should report all pregnancies, including the partners of male patients, to the Sponsor within 24 hours. The investigator should counsel the patient/partner, and discuss the risks of continuing with the pregnancy and the possible effects on the fetus. Monitoring of the patient/partner should continue until conclusion of the pregnancy. Pregnancies occurring up to 7 months after the completion of study medication must also be reported to the investigator. Please refer to Section 5.4.3 for reporting procedures.

It is not known whether trastuzumab or trastuzumab emtansine are excreted in human milk. Maternal IgG is excreted in milk and any of these monoclonal antibodies could harm infant growth and development; therefore, women should be advised to discontinue nursing during trastuzumab emtansine therapy and not to breastfeed for at least 7 months following the last dose of either study drug.

Experimental studies have reported that IgGs are present in both the pre-ejaculate and the seminal plasma. To date, there have been no clinical studies to assess the IgG profile in the pre-ejaculate and seminal plasma in male patients receiving trastuzumab or trastuzumab emtansine. Therefore, as a precaution male patients with female partners of childbearing potential are required to use highly effective form of contraception or use two forms of contraception as outlined above. Similarly, vaginal absorption of trastuzumab emtansine is unknown and therefore male patients with pregnant partners are required to use condoms for the duration of the pregnancy, and then revert to contraceptive methods as outlined above. This is to ensure that the fetus is not exposed to the study medication through vaginal absorption. In addition, sperm or blood donation should not occur for at least 7 months after the last dose of study treatment.

### 5.3 METHODS AND TIMING FOR CAPTURING AND ASSESSING SAFETY PARAMETERS

The investigator is responsible for ensuring that all AEs (see Section 5.2.1 for definition) are recorded on the AE eCRF and reported to the Sponsor in accordance with instructions provided in this section and in Sections 5.4, 5.5, and 5.6.

For each AE recorded on the AE eCRF, the investigator will make an assessment of seriousness (see Section 5.2.2, for seriousness criteria), severity (see Section 5.3.3), and causality (see Section 5.3.4).

#### 5.3.1 ADVERSE EVENT REPORTING PERIOD

Investigators will seek information on AEs at each patient contact. All AEs, whether reported by the patient or noted by study personnel, will be recorded in the patient's medical record and on the AE eCRF.

After informed consent has been obtained but prior to initiation of study drug, only SAEs caused by a protocol-mandated intervention (e.g., invasive procedures such as biopsies, discontinuation of medications) should be reported (see Section 5.4.2 for instructions for reporting SAEs).

After initiation of study treatment, all AEs, regardless of relationship to study drug, will be reported until 28 days after the last administration of study drug. After this period, the investigator is not required to actively monitor for AEs; however, the Sponsor should be notified if the investigator becomes aware of any poststudy SAEs (see Section 5.6).

### 5.3.2 ELICITING ADVERSE EVENT INFORMATION

A consistent methodology of non-directive questioning should be adopted for eliciting AE information at all patient evaluation time points. Examples of non-directive questions include the following:

"How have you felt since your last clinic visit?"

"Have you had any new or changed health problems since you were last here?"

#### 5.3.3 ASSESSMENT OF SEVERITY OF ADVERSE EVENTS

The AE grading (severity) scale found in the NCI CTCAE (v. 4.0) will be used for assessing AE severity (see Table 6).

Table 6 Adverse Event Severity Grading Scale

| | Severity | Alternate Description a |
|---|---|---|
| Grade | | |
| 1 | Mild (apply event-specific NCI CTCAE grading criteria) | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate (apply event-specific NCI CTCAE grading criteria) | Minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental ADL <sup>b</sup> |
| 3 | Severe (apply event-specific NCI CTCAE grading criteria) | Severe or medically significant but<br>not immediately life-threatening; hospitalization<br>or prolongation of hospitalization indicated;<br>disabling; limiting self-care ADL° |
| 4 | Very severe, life-threatening,<br>or disabling (apply event-specific<br>NCI CTCAE grading criteria) | Life-threatening consequences; urgent intervention indicated |
| 5 | Death related to AE | |

ADL = activities of daily living; AE = adverse event; CTCAE = Common Terminology Criteria for Adverse Events; NCI = National Cancer Institute.

The NCI CTCAE v4.0 can be found at:

http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm#ctc\_40 Note: Regardless of severity, some events may also meet regulatory seriousness criteria. Refer to definition of a serious AE (see Section 5.2.2).

- <sup>a</sup> Use these alternative definitions for Grade 1, 2, 3, and 4 events when the observed or reported AE is not in the NCI CTCAE listing.
- b Instrumental ADL refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
- Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

#### 5.3.4 ASSESSMENT OF CAUSALITY OF ADVERSE EVENTS

Investigators should use their knowledge of the patient, the circumstances surrounding the event, and an evaluation of any potential alternative causes to determine whether or not an AE is considered to be related to study drugs, indicating "yes" or "no" accordingly. To ensure consistency of causality assessments, investigators should apply the general guidelines outlined in Table 7.

#### Table 7 Guidance for Causal Attribution of Adverse Event/Serious Adverse Event

Is the AE/SAE suspected to be caused by the investigational product based on facts, evidence, science-based rationales, and clinical judgment?

YES There is a plausible temporal relationship between the onset of the AE and administration of the investigational product, and the AE cannot be readily explained by the patient's clinical state, intercurrent illness, or concomitant therapies; and/or the AE follows a known pattern of response to the investigational product; and/or the AE abates or resolves upon discontinuation of the investigational product or dose reduction and, if applicable, reappears upon re-challenge.

Investigators should apply facts, evidence, or rationales based on scientific principles and clinical judgment to support a causal/contributory association with an investigational product.

#### NO <u>AEs will be considered related, unless they fulfill the criteria as specified below.</u>

Evidence exists that the AE has an etiology other than the investigational product (e.g., pre-existing medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the AE has no plausible temporal relationship to administration of the investigational product (e.g., cancer diagnosed 2 days after first dose of study drug).

Note: The investigator's assessment of causality for individual AE reports is part of the study documentation process. Regardless of the "Yes" or "No" causality assessment for individual AE reports, the Sponsor will promptly evaluate all reported SAEs against cumulative product experience to identify and expeditiously communicate possible new safety findings to investigators and applicable regulatory authorities. <a href="Attribution of SAEs will be reviewed on an ongoing basis">Attribution of SAEs will be reviewed on an ongoing basis</a>, and may be changed as additional clinical data emerges (e.g., reversibility of AE, new clinical findings in patient with AE, effects of retreatment, AEs in other patients).

In addition to assessing causality with respect to study drugs, investigators should also assess whether other factors (e.g., disease under study, concurrent illness, concomitant medication, or study procedure) may have caused the event, using similar guidance.

The investigator's assessment of causality for individual AE reports is part of the study documentation process. Regardless of the "Yes" or "No" causality assessment for individual AE reports, the Sponsor will promptly evaluate all reported serious AEs against cumulative product experience to identify and expeditiously communicate possible new safety findings to investigators and applicable regulatory authorities.

For patients receiving combination therapy, causality will be assessed individually for each protocol-mandated therapy.

#### 5.3.5 PROCEDURES FOR RECORDING ADVERSE EVENTS

Investigators should use correct medical terminology/concepts when recording AEs on the AE eCRF. Avoid colloquialisms and abbreviations.

There is one eCRF page for recording AEs or SAEs.

Only one AE term should be recorded in the event field on the AE eCRF.

#### 5.3.5.1 Diagnosis *versus* Signs and Symptoms

#### Infusion-related Reactions

AEs that occur during or within 24 hours after study drug infusion should be captured as individual signs and symptoms rather than a diagnosis of allergic reaction or infusion-related reaction. However, a diagnosis has to be captured as an AE if signs and symptoms constitute a diagnosis of allergic reaction/hypersensitivity or infusion-related reaction and are classified as SAEs; all such symptoms have to be described in the narrative (e.g., in the Additional Case Details field of the eCRF).

#### **Other Adverse Events**

For AEs other than infusion-related reactions, a diagnosis (if known) should be recorded on the AE eCRF rather than individual signs and symptoms (e.g., record only liver failure or hepatitis rather than jaundice, asterixis, and elevated transaminases). However, if a constellation of signs and/or symptoms cannot be medically characterized as a single diagnosis or syndrome at the time of reporting, each individual event should be recorded on the AE eCRF. If a diagnosis is subsequently established, all previously reported AEs based on signs and symptoms should be nullified and replaced by one AE report based on the single diagnosis, with a starting date that corresponds to the starting date of the first symptom of the eventual diagnosis.

#### 5.3.5.2 Adverse Events Occurring Secondary to Other Events

In general, AEs occurring secondary to other events (e.g., cascade events or clinical sequelae) should be identified by their primary cause. For example, if severe diarrhea is known to have resulted in dehydration, it is sufficient to record only diarrhea as an AE or SAE on the eCRF.

However, medically significant AEs occurring secondary to an initiating event that are separated in time should be recorded as independent events on the eCRF. For example, if a severe gastrointestinal hemorrhage leads to renal failure, both events should be recorded separately on the eCRF.

#### 5.3.5.3 Persistent or Recurrent Adverse Events

A persistent AE is one that extends continuously, without resolution, between patient evaluation time points. Such events should only be recorded once on the AE eCRF. The initial severity of the event should be recorded, and the severity should be updated to reflect the most extreme severity any time the event worsens. If the event becomes serious, the AE eCRF should be updated to reflect this.

A recurrent AE is one that resolves between patient evaluation time points and subsequently recurs. Each recurrence of an AE should be recorded separately on the AE eCRF.

#### 5.3.5.4 Abnormal Laboratory Values

Only clinically significant laboratory abnormalities that require active management will be recorded as AEs or SAEs on the eCRF (e.g., abnormalities that require study drug dose modification, discontinuation of study treatment, more frequent follow-up assessments, further diagnostic investigation, etc.).

If the clinically significant laboratory abnormality is a sign of a disease or syndrome (e.g., alkaline phosphatase and bilirubin 5 × ULN of normal associated with cholecystitis), only the diagnosis (e.g., cholecystitis) needs to be recorded on the AE eCRF.

If the clinically significant laboratory abnormality is not a sign of a disease or syndrome, the abnormality itself should be recorded as an AE or SAE on the eCRF. If the laboratory abnormality can be characterized by a precise clinical term, the clinical term should be recorded as the AE or SAE. For example, an elevated serum potassium level of 7.0 mEq/L should be recorded as "hyperkalemia."

Observations of the same clinically significant laboratory abnormality from visit to visit should not be repeatedly recorded as AEs or SAEs on the eCRF, unless their severity, seriousness, or etiology changes.

#### 5.3.5.5 Deaths

Deaths that occur during the protocol-specified AE reporting period (see Section 5.3.1), that are attributed by the investigator solely to progression of mBC or mGC should be recorded only on the Study Completion/Early Discontinuation eCRF. All other on-study deaths, regardless of relationship to study drug, must be recorded on the AE eCRF and immediately reported to the Sponsor (see Section 5.4.2). The IDMC will monitor the frequency of death from all causes.

Death should be considered an outcome and not a distinct event. The event or condition that caused or contributed to the fatal outcome should be recorded as the single medical concept on the AE eCRF. Generally, only one such event should be reported. If the cause of death is unknown and cannot be ascertained at the time of reporting, "unexplained death" should be recorded on the AE eCRF. If the cause of death later becomes available (e.g., after autopsy), "unexplained death" should be replaced by the established cause of death.

During post-study survival follow-up, deaths attributed to progression of mBC or LA/mGC should be recorded only on the Survival eCRF.

#### 5.3.5.6 Pre-Existing Medical Conditions

A pre-existing medical condition is one that is present at the start of this study. Such conditions should be recorded on the Medical and Surgical History eCRF.

A pre-existing medical condition should be recorded as an AE <u>only</u> if the frequency, severity, or character of the condition worsens during the study. When recording such events on the AE eCRF, it is important to convey the concept that the pre-existing condition has changed by including applicable descriptors (e.g., "more frequent headaches").

#### 5.3.5.7 Lack of Efficacy or Clinical Worsening

Events that are clearly consistent with the expected pattern of progression of mBC or LA/mGC should not be recorded as AEs. These data will be captured as efficacy assessment data only. In most cases, the expected pattern of progression will be based on the RECIST criteria. In rare cases, the determination of clinical progression will be based on symptomatic deterioration. However, every effort should be made to document progression using objective criteria. If there is any uncertainty as to whether an event is due to PD, it should be reported as an AE.

#### 5.3.5.8 Hospitalization or Prolonged Hospitalization

Any AE that results in hospitalization or prolonged hospitalization should be documented and reported as a SAE unless specifically instructed otherwise in this protocol.

There are some hospitalization scenarios that do not require reporting as an SAE when there is no occurrence of an AE. These scenarios include a planned hospitalization or prolonged hospitalization to:

- Perform an efficacy measurement for the study
- Undergo a diagnostic or elective surgical procedure for a pre-existing medical condition that has not changed
- Receive scheduled therapy for the target disease of the study

### 5.4 IMMEDIATE REPORTING REQUIREMENTS FROM INVESTIGATOR TO THE SPONSOR

Certain events require immediate reporting to allow the Sponsor to take appropriate measures to address potential new risks in a clinical trial. The investigator must report such events to the Sponsor immediately; under no circumstances should reporting take place more than 24 hours after the investigator learns of the event. The following is a list of events that the investigator must report to the Sponsor within 24 hours after learning of the event, regardless of relationship to study drug:

- SAEs
- Non-serious AESIs
- Pregnancies

The investigator must report new significant follow-up information for these events to the Sponsor immediately (i.e., no more than 24 hours) after becoming aware of the information. New significant information includes the following:

- New signs or symptoms or a change in the diagnosis
- Significant new diagnostic test results
- Change in causality based on new information
- Change in the event's outcome, including recovery
- Additional narrative information on the clinical course of the event

Investigators must also comply with local requirements for reporting SAEs to the local health authority and Institutional Review Board/Ethics Committee (IRB/EC).

#### 5.4.1 EMERGENCY MEDICAL CONTACTS

### MEDICAL MONITOR (SPONSOR'S MEDICAL RESPONSIBLE) CONTACT INFORMATION

To ensure the safety of study patients, an Emergency Medical Call Center Help Desk will access the Sponsor Medical Emergency List, escalate emergency medical calls, provide medical translation service (if necessary), connect the investigator with a Sponsor Medical Monitor, and track all calls. The Emergency Medical Call Center Help Desk will be available 24 hours per day, 7 days per week. Toll-free numbers for the Help Desk and Medical Monitor contact information will be distributed to all investigators (see "Protocol Administrative and Contact Information and List of Investigators").

# 5.4.2 REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS AND NON-SERIOUS ADVERSE EVENTS OF SPECIAL INTEREST

For reports of SAEs and non-serious AESIs, investigators should record all case details that can be gathered immediately (i.e., no more than 24 hours) on the AE eCRF and submit the report via the electronic data capture (EDC) system. A report will be generated and sent to the Sponsor Safety Risk Management by the EDC system.

In the event that the EDC system is unavailable, a paper SAE/Non-Serious AE of Special Interest CRF and Fax Coversheet should be completed and faxed to the Sponsor Safety Risk Management or its designee immediately (i.e., no more than 24 hours) after learning of the event, using the fax numbers provided to investigators (see "Protocol Administrative and Contact Information & List of Investigators"). Once the EDC system is available, all information will need to be entered and submitted via the EDC system.

#### 5.4.3 REPORTING REQUIREMENTS FOR PREGNANCIES

#### **5.4.3.1** Pregnancies in Female Patients

Female patients of childbearing potential will be instructed to immediately inform the investigator if they become pregnant during the study or within 7 months after the last dose of study drug. A Pregnancy Report eCRF should be completed by the investigator immediately (i.e., no more than 24 hours)

after learning of the pregnancy and submitted via the EDC system. A Pregnancy Report will automatically be generated and sent to the Sponsor Safety Risk Management. Pregnancy should not be recorded on the AE eCRF. The investigator should have the patient discontinue the study drug and discuss with the patient the risks of the pregnancy and the possible effects on the fetus. Monitoring of the patient should continue until conclusion of the pregnancy.

In the event that the EDC system is unavailable, a Pregnancy Report worksheet and Pregnancy Fax Coversheet should be completed and faxed to the Sponsor Safety Risk Management or its designee immediately (i.e., no more than 24 hours) after learning of the pregnancy, using the fax numbers provided to investigators (see "Protocol Administrative and Contact Information & List of Investigators").

#### 5.4.3.2 Pregnancies in Female Partners of Male Patients

Male patients will be instructed through the Informed Consent Form to immediately inform the investigator if their partner becomes pregnant during the study or within 7 months after the last dose of study drug. A Pregnancy Report eCRF should be completed by the investigator immediately (i.e., no more than 24 hours) after learning of the pregnancy and submitted via the EDC system. Attempts should be made to collect and report details of the course and outcome of any pregnancy in the partner of a male patient exposed to study drug. The pregnant partner will need to sign an Authorization for Use and Disclosure of Pregnancy Health Information to allow for follow-up on her pregnancy. Once the authorization has been signed, the investigator will update the Pregnancy Report eCRF with additional information on the course and outcome of the pregnancy. An investigator who is contacted by the male patient or his pregnant partner may provide information on the risks of the pregnancy and the possible effects on the fetus, to support an informed decision in cooperation with the treating physician and/or obstetrician.

In the event that the EDC system is unavailable, follow reporting instructions provided in Section 5.4.3.1.

#### 5.4.3.3 Abortions

Any spontaneous abortion should be classified as an SAE (as the Sponsor considers spontaneous abortions to be medically significant events), recorded on the AE eCRF, and reported to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2).

#### 5.4.3.4 Congenital Anomalies/Birth Defects

Any congenital anomaly/birth defect in a child born to a female patient or female partner of a male patient exposed to study drug should be classified as an SAE, recorded on the AE eCRF, and reported to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2).

### 5.5 FOLLOW-UP OF PATIENTS AFTER ADVERSE EVENTS

#### 5.5.1 INVESTIGATOR FOLLOW-UP

The investigator should follow all unresolved AEs and until the events are resolved or stabilized, the patient is lost to follow-up, or it has been determined that the study treatment or participation is not the cause of the AE/SAE. Resolution of AEs and SAEs (with dates) should be documented on the AE eCRF and in the patient's medical record to facilitate source data verification (SDV).

All pregnancies reported during the study should be followed until pregnancy outcome. If the EDC system is not available at the time of pregnancy outcome, follow reporting instructions provided in Section 5.4.3.1.

#### 5.5.2 Sponsor Follow-up

For SAEs, non-serious AESIs, and pregnancies, the Sponsor or a designee may follow-up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details and outcome information (e.g., from hospital discharge summaries, consultant reports, autopsy reports) in order to perform an independent medical assessment of the reported case.

#### 5.6 POST-STUDY ADVERSE EVENTS

At the time of study completion or study discontinuation, the investigator should instruct each patient to report to the investigator any subsequent AEs that the patient's physician believes could be related to prior study drug treatment or study procedures.

The investigator is not required to actively monitor patients for AEs after the end of the AE reporting period (defined as 28 days after the last dose of study drug). However, the Sponsor should be notified if the investigator becomes aware of any death or other SAE occurring after the end of the AE reporting period, regardless of causality.

The investigator should report these events directly to Roche Safety Risk Management via telephone or via facsimile using the Roche Clinical Trial (SAE) Reporting Form.

# 5.7 EXPEDITED REPORTING TO HEALTH AUTHORITIES, INVESTIGATORS, INSTITUTIONAL REVIEW BOARDS, AND ETHICS COMMITTEES

To determine reporting requirements for single AE cases, the Sponsor will assess the expectedness of these events using the following reference documents:

Trastuzumab emtansine and capecitabine Investigator's Brochures

The Sponsor will compare the severity of each event and the cumulative event frequency reported for the study with the severity and frequency reported in the applicable reference document.

Reporting requirements will also be based on the investigator's assessment of causality and seriousness, with allowance for upgrading by the Sponsor as needed.

The IDMC will closely monitor the incidence of these expected events during the study. An aggregate report of any clinically relevant imbalances that do not favor the test product will be submitted to health authorities.

### 6. <u>STATISTICAL CONSIDERATIONS AND ANALYSIS</u> PLAN

The design of this study includes: Phase I, Randomized Phase II and different cohorts. Corresponding analyses as described in the protocol will be performed when all data for a particular cohort and study phase are collected and cleaned.

#### Phase I: Patients with mBC:

Enrollment into Cohort 1, patients with HER2-positive mBC, will open first. Enrolled patients will receive study drug until Investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

Patients randomized in Phase II will receive study drug until investigatorassessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.

The primary analysis of BOR will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever comes first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after the randomization of the first patient.

The EOS analysis will include an updated analysis of BOR, which will be done in a purely exploratory manner.

#### Phase I: Patients with mGC:

Once the MTD is established for Cohort 1, enrollment of patients with HER2-positive and LA/mGC into Cohort 2 will be opened.

Enrolled patients will receive study drug until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.

#### 6.1 DETERMINATION OF SAMPLE SIZE

#### Sample Size for Phase I: mBC

This part will be based on a classical 3 plus 3 Phase I design. A minimum of 6 and up to 18 patients will be enrolled into Cohort 1. There is no formal sample size estimation for this part.

### Sample Size for Randomized Phase II: Exploration of Efficacy and Safety in mBC

The sample size for the primary endpoint BOR is based on a Fisher's exact test with an alpha level of 5% (one-sided),<sup>48,49</sup> power of 80% and the clinical assumption of a BOR rate of 43% with trastuzumab emtansine alone and 62.5% with the combination of trastuzumab emtansine and capecitabine. Approximately 210 patients (105 patients in each treatment group), including a 15% withdrawal rate, will be randomized with a 1:1 ratio to trastuzumab emtansine alone or the combination of trastuzumab emtansine and capecitabine.

An expected BOR rate of 43.6% (95% CI: 38.6%–48.6%) for patients receiving trastuzumab emtansine alone was chosen based on previously published data for T-DM1 in patients with unresectable, locally advanced or mBC previously treated with a taxane and trastuzumab (EMILIA study).<sup>27</sup>

The BOR rates for patients treated with the combination of T-DM1 and capecitabine were chosen based on recent results from other combination studies of T-DM1 plus chemotherapy or trastuzumab plus capecitabine. Response rates were based on those observed in patients with HER2-positive mBC in a Phase Ib/IIa study (BP22752) that compared the combination of trastuzumab emtansine with docetaxel, with or without pertuzumab (ORR: 76% [95% CI: 53%–92%]), and also in a Phase II study that compared the combination of trastuzumab with docetaxel, with or without capecitabine (ORRs: 72.7% [95% CI: 63.4%–80.8%] and 70.5% [95% CI: 61.2%–78.8%]).<sup>41</sup>

Increased BOR rates for the combination treatment compared with single-agent trastuzumab emtansine are in line with previously published results of a randomized Phase III study in patients with locally advanced or mBC treated with the combination of trastuzumab with capecitabine *versus* capecitabine alone (ORR: 48.1% *versus* 27.0%, odds ratio = 2.50, p = 0.0115).9

The estimation of sample size was performed by Nquery<sup>®</sup> and EAST<sup>®</sup> programs.

#### **Stratification Factors**

The following stratification factor will be implemented in the Randomized Phase II of the study:

• Number of prior lines of treatment for metastatic disease (≤1 or >1; excluding single-agent hormones)

A treatment line is any regimen given to a patient from treatment initiation until confirmed PD.

#### Sample Size for Phase I: mGC

This part will be based on a classical 3 plus 3 Phase I design. From 3 to 12 patients might be enrolled into Cohort 2. There is no formal sample size estimation for this part.

#### 6.2 SUMMARIES OF CONDUCT OF STUDY

#### Phase I: Patients with mBC

Due to the small sample size, per-protocol (PP) population will not be defined for the Phase I, Cohort 1.

Major protocol violations will be summarized by treatment dosage. Median follow-up will be estimated for Phase I, Cohort 1.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

For the Randomized Phase II part of the study, a PP population will be defined (Section 6.4).

Patient enrollment, duration of follow-up, discontinuation from study treatment and study, and reasons for study discontinuation will be summarized by treatment group for all randomized patients. In addition, major protocol violations will be summarized by treatment arm.

#### Phase I: Patients with LA/mGC

Due to the small sample size, a PP population will not be defined for the Phase I, Cohort 2.

Major protocol violations will be summarized by treatment dosage. Median follow-up will be estimated for Phase I, Cohort 2.

### 6.3 SUMMARIES OF TREATMENT GROUP COMPARABILITY

#### Phase I: mBC

As Phase I is the MTD-Finding part of the study, there are no treatment group comparisons for this part of the study.

Demographics, medical history, and baseline characteristics will be summarized. Continuous variables will be summarized using median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range. Categorical variables will be summarized by the number and percentage of patients for each treatment dosage.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

The Randomized Phase II part of the study is designed to explore the efficacy and safety of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone.

Demographics, medical history, and baseline characteristics will be summarized. Continuous variables will be summarized using median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range. Categorical variables will be summarized by the number and percentage of patients for each treatment group.

#### Phase I: mGC

As Phase I is the MTD-Finding part of the study, there are no treatment group comparisons for this part of the study.

Demographics, medical history and baseline characteristics will be summarized. Continuous variables will be summarized using median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range. Categorical variables will be summarized by the number and percentage for each treatment dosage.

#### 6.4 EFFICACY ANALYSES

#### Phase I, Cohort 1: mBC

The main analysis population will be the DLT-evaluable population as defined in Section 6.5.

#### Randomized Phase II: Exploration of Efficacy in mBC

The main analysis population for the efficacy analysis will be the intent-to-treat population (ITT), which will include all patients in the Randomized Phase II part of the study. The PP population will include all ITT patients who have at least one post-baseline tumor assessment during the Phase II part and no major protocol violations, which will be defined in the statistical analysis plan (SAP).

#### Phase I, Cohort 2: mGC

The main analysis population will be the DLT-evaluable population as defined in Section 6.5.

#### 6.4.1 PRIMARY EFFICACY ENDPOINT

#### Phase I. Cohort 1: Patients with mBC

The primary objectives are defining the MTD and establishing the safety profile. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination.

ORR, as a main efficacy endpoint, will be assessed via BOR rate. The BOR is defined as the best response recorded from the date of enrollment until PD,

death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

#### Randomized Phase II: Exploration of Efficacy in mBC

The primary efficacy endpoint for the Randomized Phase II part of the study is the ORR as assessed via BOR. The BOR is defined as the best response recorded from the start or randomization into the Phase II part of the study and until PD, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. To be assigned a status of PR or CR, i.e., to be a responder, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 28 days after the criteria for response are first met, i.e., patients need to have two consecutive assessments of PR or CR.

The primary hypothesis of interest when comparing ORR – as assessed via BOR – between the two treatment groups (combination of trastuzumab emtansine and capecitabine *versus* trastuzumab emtansine alone) is:

- H0: π TDM1 = π trastuzumab emtansine + capecitabine Where π trastuzumab emtansine is BOR in TDM1 and π trastuzumab emtansine + capecitabine is BOR in trastuzumab emtansine + capecitabine
- H1:  $\pi$  trastuzumab emtansine  $\neq \pi$  trastuzumab emtansine + capecitabine

The number and proportions of responders and non-responders (based on BOR) together with 90% Clopper-Pearson Cls will be presented for each treatment group.

The difference in BOR between treatment groups will be displayed with associated 90% CIs using the Hauck-Anderson approach and p-values for the Fisher's exact test.

Logistic analysis will be used to assess the influence of the stratification factor and baseline covariates in an exploratory manner.

The primary analysis of BOR will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever comes first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after the randomization of the first patient.

#### Phase I, Cohort 2: Patients with LA/mGC

The primary objectives are defining the MTD and establishing the safety profile. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination.

ORR, as a main efficacy endpoint, will be assessed via BOR rate. The BOR is defined as the best response recorded from the date of enrollment until PD, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

#### 6.4.2 SECONDARY EFFICACY ENDPOINTS

#### Phase I, Cohort 1: mBC

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### Randomized Phase II: Exploration of Efficacy in mBC

The secondary efficacy endpoints for the Randomized Phase II will be:

- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

TTR is defined as the time from randomization to first documentation of confirmed PR or CR (whichever occurs first). Patients who do not have a confirmed response will be censored at the date of the last tumor assessment.

DoR is defined as the period from the date of first recorded PR or CR until the date of PD or death from any cause. Patients with no documented progression after CR or PR will be censored at the last date at which they are known to have had the CR or PR. The method for handling censoring is the same as described for PFS below. Only patients with a BOR of CR or PR (i.e., responders) will be included in the analysis of DoR.

For patients with a BOR of CR or PR, TTR is defined as the time from randomization to the date of first CR or PR. The censoring rules will be similar to those of the PFS.

TTP is defined as time from randomization to the first occurrence of PD. Patients who have not progressed at the time of study completion (including patients who have died before PD) or who are lost to follow-up are censored at the date of the last tumor assessment.

TTF is defined as time from randomization until treatment failure, i.e., to PD, death, withdrawal due to AE or laboratory abnormality, or refusal of treatment. Patients who do not experience any of the above events while on study will be censored on the day of their last tumor assessment.

PFS is defined as the time from randomization until the first documented progression of disease or death from any cause, whichever occurs first. Patients with no PFS events will be censored at the time of the last evaluable tumor assessment. Patients with no post-baseline tumor assessment will be censored at the time of randomization plus 1 day.

OS is defined as the time from randomization until the date of death, regardless of the cause of death. Patients who are alive at the time of data cut-off will be censored at the date of the last follow-up assessment.

Estimates for the survivor function of both treatment groups for TTR, DoR, TTP, TTF, and OS will be obtained by using the Kaplan-Meier method. HRs and associated 90% CIs will be estimated from non-stratified and stratified (based on the stratification factor) Cox regression models.

CBR includes patients whose best (confirmed) response was PR, CR or SD that lasted at least 6 months. CBR will be summarized in a similar way to the primary efficacy endpoint, ORR as assessed by BOR.

#### Phase I, Cohort 2: mGC

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### 6.5 SAFETY ANALYSES

#### Safety Population Phase I, Cohort 1: mBC

The DLT-evaluable population is defined as all enrolled and treated patients who have not experienced any major protocol violation (including violation of the inclusion and exclusion criteria) and completed Cycle 1.

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

The safety population (SP) will include all patients who received at least one dose of study medication during Phase I. Safety endpoints will be summarized by treatment dosage.

Safety parameters for this part of the study will be summarized by treatment dose. The summaries of AEs, SAEs, AEs that caused discontinuation from the study treatment and/or study, and AESIs will be analyzed in a similar way to AEs in Phase II.

The incidence of AEs and SAEs will be summarized according to the primary SOC and, within each SOC, by MedDRA preferred term. Based on the safety profile of trastuzumab emtansine, time to onset of the first episode of any AESI described in Section 5 will also be summarized via Kaplan-Meier estimates. Additional summaries by frequency tables will also be provided for the AESIs. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry will be presented in shift tables of NCI-CTC grade at baseline *versus* worst grade during treatment for Phase I, Cohort 2, and overall.

LVEF will be summarized over time using mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### Randomized Phase II: Exploration of Safety in mBC

The SP will include all patients who received at least one dose of study medication during the Randomized Phase II part of the study. Safety endpoints will be summarized by treatment group.

Safety endpoints during Phase II will be assessed via total AEs, Grade ≥3 AEs, SAEs, AESIs (as described in Section 5), fatal AEs and their causes, events to monitor, premature withdrawal from study medication and/or study, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by the Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Based on the safety profile of trastuzumab emtansine, time to onset of the first episode of any AESI described in Section 5 will also be summarized via Kaplan-Meier estimates. Additional summaries by frequency tables will be provided for the AESIs. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology, and biochemistry will be presented in shift tables of NCI-CTCAE grade at baseline *versus* worst grade during treatment for the Randomized Phase II part of the study.

LVEF will be summarized over time using mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations, will be analyzed in a similar way. The exposure to study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### Safety Population Phase I, Cohort 2: LA/mGC

The DLT-evaluable population is defined as all enrolled and treated patients who have not experienced any major protocol violation (including violation of the inclusion and exclusion criteria) and have completed Cycle 1.

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

The SP will include all patients who received at least one dose of study medication during Phase I. Safety endpoints will be summarized by treatment dosage.

Safety parameters will be analyzed in a similar way to safety parameters in Phase I, Cohort 1: mBC.

#### 6.6 PHARMACODYNAMIC ANALYSES

No pharmacodynamic analyses are planned for this study.

#### 6.7 PHARMACOKINETIC ANALYSES

#### For Phase I only (Patients with mBC and LA/mGC):

The following PK parameters of trastuzumab emtansine, capecitabine and their metabolites (including but not limited to those listed below) will be determined only in the Phase I part of the study for Cohort 1 and Cohort 2 in all patients who receive study treatment using either non-compartmental and/or population methods, if data allow:

- Serum concentrations of trastuzumab emtansine (conjugate) and total trastuzumab
- Plasma concentrations of DM1, capecitabine and its active metabolite 5-FU
- Total exposure (e.g., AUC)
- Cmax
- CL
- V<sub>d</sub>
- T<sub>1/2</sub>

The PK of trastuzumab emtansine, total trastuzumab and DM1 will be compared with historical single-agent PK data to evaluate the potential effect of capecitabine on the PK of trastuzumab emtansine and related analytes. The PK of capecitabine and its active metabolite 5-FU in Cycle 1 (in the absence of trastuzumab emtansine) will be compared with the PK of Cycle 2 (in the presence of trastuzumab emtansine) to evaluate the potential effect of trastuzumab emtansine on the PK of capecitabine and 5-FU.

All PK parameters will be listed and tabulated by treatment dose and by Cohort. Descriptive summary statistics including arithmetic mean, geometric mean (e.g., AUC and  $C_{max}$ ), median, range, s.d., and coefficient of variation will be presented for each cohort. Nonlinear mixed effects modeling will also be used; details will be presented in the SAP.

PK samples can be obtained ad hoc in case of a SAE or unexpected toxicities which may suggest a potential drug-drug interaction.

#### 6.8 EXPLORATORY ANALYSES

For all patients with mBC (Phase I, cohort 1; Phase II Exploration of Efficacy and Safety in mBC), a retrospective central confirmation of the HER2 status will be done. Further exploratory analysis for HER2-positive patients (based on central confirmation) will be done for selected endpoints such as BOR and safety endpoints (AEs, SAEs, Grade ≥ 3 AEs, and AESIs).

### For the Randomized Phase II only: Exploration of Efficacy and Safety in Patients with mBC:

Subgroup analysis for BOR, safety endpoints (AEs, SAEs, Grade  $\geq$  3 AEs, and AESIs) in Phase II will be presented for: elderly *versus* younger patients, patients with ECOG 0–1 *versus* ECOG 2, and patients with  $\leq$  versus >1 prior treatment regimen for metastatic disease.

More details about subgroups will be provided in the SAP.

#### **Pharmacoeconomic Endpoint:**

The resource expenditure due to hospitalizations that are not study-defined evaluations while on study treatment will be evaluated. The number of hospital visits, number of days admitted, and type of visits (emergency department *versus* inpatient care) will be collected. The reason for admission (PD *versus* AE) will also be assessed.

#### 6.9 INTERIM ANALYSES

There is no formal efficacy interim analysis.

However, an IDMC will recommend whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 25, 75, and 150 patients have received at least 3 cycles (Cycle 3 Day 1) of treatment in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the course of the Randomized Phase II of the study or as requested.

Efficacy data will be provided only if required by the IDMC to estimate the risk-benefit balance for the patients. Further details on the function and logistics of the IDMC will be provided in the IDMC Charter.

#### 7. DATA COLLECTION AND MANAGEMENT

#### 7.1 DATA QUALITY ASSURANCE

The Sponsor will be responsible for data management of this study, including quality checking of the data. Data entered manually will be collected via EDC using eCRFs. The sites will be responsible for data entry into the EDC system. In the event of discrepant data, the Sponsor will request data clarification from the sites, which the sites will resolve electronically in the EDC system.

The Sponsor will produce an EDC Study Specification document that describes the quality checking to be performed on the data. Central laboratory data and other electronic data will be sent directly to the Sponsor, using the Sponsor's standard procedures to handle and process the electronic transfer of these data.

eCRFs and correction documentation will be maintained in the EDC system's audit trail. System backups for data stored by the Sponsor and records retention for the study data will be consistent with the Sponsor's standard procedures.

#### 7.2 ELECTRONIC CASE REPORT FORMS

eCRFs are to be completed using a Sponsor-designated EDC system. Sites will receive training and have access to a manual for appropriate eCRF completion. eCRFs will be submitted electronically to the Sponsor and should be handled in accordance with instructions from the Sponsor.

All eCRFs should be completed by designated, trained site staff. eCRFs should be reviewed and electronically signed and dated by the investigator or a designee.

At the end of the study, the investigator will receive patient data for his or her site in a readable format on a compact disc that must be kept with the study records. Acknowledgment of receipt of the compact disc is required.

#### 7.3 SOURCE DATA DOCUMENTATION

Study monitors will perform ongoing SDV to confirm that critical protocol data (i.e., source data) entered into the eCRFs by authorized site personnel are accurate, complete, and verifiable from source documents.

Source documents (paper or electronic) are those in which patient data are recorded and documented for the first time. They include, but are not limited to, hospital records, clinical and office charts, laboratory notes, memoranda, patient-reported outcomes, evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies of transcriptions that are certified after verification as being accurate and complete, microfiche, photographic negatives, microfilm or magnetic media, X-rays, patient files, and records kept at pharmacies, laboratories, and medico-technical departments involved in a clinical trial.

Source documents that are required to verify the validity and completeness of data entered into the eCRFs must not be obliterated or destroyed.

To facilitate SDV, the investigators and institutions must provide the Sponsor with direct access to applicable source documents and reports for trial-related monitoring, Sponsor audits, and IRB/EC review. The investigational site must also allow inspection by applicable health authorities.

#### 7.4 USE OF COMPUTERIZED SYSTEMS

When clinical observations are entered directly into an investigational site's computerized medical record system (i.e., in lieu of original hardcopy records), the electronic record can serve as the source document if the system has been validated in accordance with health authority requirements pertaining to computerized systems used in clinical research. An acceptable computerized data collection system (for clinical research purposes) would be one that (1) allows data entry only by authorized individuals; (2) prevents the deletion or alteration of previously entered data and provides an audit trail for such data changes (e.g., modification of file); (3) protects the database from tampering; and (4) ensures data preservation.

In collaboration with the study monitor, Sponsor's Quality Assurance group may assist in assessing whether electronic records generated from computerized medical record systems used at investigational sites can serve as source documents for the purposes of this protocol.

If a site's computerized medical record system is not adequately validated for the purposes of clinical research (as opposed to general clinical practice), applicable hardcopy source documents must be maintained to ensure that critical protocol data entered into the eCRFs can be verified.

#### 7.5 RETENTION OF RECORDS

U.S. FDA regulations (21 Code of Federal Regulations §312.62[c]) and the ICH Guideline for Good Clinical Practice (GCP) (see Section 4.9 of the guideline) require that records and documents pertaining to the conduct of this study and the distribution of investigational drug, including eCRFs, Consent Forms, laboratory test results, and medication inventory records, must be retained by the Principal Investigator for 2 years after the last marketing application approval in an ICH region or after at least 2 years have elapsed since formal discontinuation of clinical development of the investigational product. All state and local laws for retention of records also apply.

No records should be disposed of without the written approval of the Sponsor. Written notification should be provided to the Sponsor for transfer of any records to another party or moving them to another location.

For studies conducted outside the United States under a U.S. Investigational New Drug (IND) application, the Principal Investigator must comply with the record retention requirements set forth in the U.S. FDA IND regulations and the relevant national and local health authorities, whichever is longer.

### 8. ETHICAL CONSIDERATIONS

#### 8.1 COMPLIANCE WITH LAWS AND REGULATIONS

This study will be conducted in full conformance with the ICH E6 guideline for GCP and the principles of the Declaration of Helsinki, or the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual. The study will comply with the requirements of the ICH E2A guideline (Clinical Safety Data Management: Definitions and Standards for Expedited Reporting). Studies conducted in the United States or under a U.S. IND application will comply with U.S. FDA regulations and applicable local, state, and federal laws. Studies conducted in the European Union (EU)/European economic area (EEA) will comply with the EU Clinical Trial Directive (2001/20/EC).

#### 8.2 INFORMED CONSENT

Sponsor's Sample Informed Consent Form will be provided to each site. If applicable, it will be provided in a certified translation of the local language. The Sponsor or its designee must review and approve any proposed deviations from the Sample Informed Consent Form or any alternate Consent Forms proposed by the site before IRB/EC submission. The final IRB/EC-approved Consent Forms must be provided to the Sponsor for health authority submission purposes according to local requirements.

The Consent Form must be signed and dated by the patient or the patient's legally authorized representative before his or her participation in the study. The case history or clinical records for each patient shall document the informed consent process and that written informed consent was obtained prior to participation in the study.

A copy of each signed Consent Form must be provided to the patient or the patient's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

All signed and dated Consent Forms must remain in each patient's study file and must be available for verification by study monitors at any time.

The Informed Consent Form should be revised whenever there are changes to procedures outlined in the informed consent or when new information becomes available that may affect the willingness of the patient to participate.

For any updated or revised Consent Forms, the case history for each patient shall document the informed consent process and that written informed consent was obtained for the updated/revised Consent Form for continued participation in the study. The final revised IRB/EC-approved Informed Consent Form must be provided to the Sponsor for regulatory purposes.

If the site uses a separate Authorization Form for patient authorization to use and disclose personal health information under the U.S. Health Insurance Portability and Accountability Act (HIPAA) regulations, the review, approval,

and other processes outlined above apply except that IRB/IEC review and approval may not be required per study site policies.

### 8.3 INSTITUTIONAL REVIEW BOARD OR ETHICS COMMITTEE

This protocol, the Informed Consent Forms, any information to be given to the patient, and relevant supporting information must be submitted to the IRB/EC by the Principal Investigator and reviewed and approved by the IRB/EC before the study is initiated. In addition, any patient enrollment materials must be approved by the IRB/EC.

The Principal Investigator is responsible for providing written summaries of the status of the study to the IRB/EC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC. Investigators are also responsible for promptly informing the IRB/EC of any protocol amendments.

In addition to the requirements to report protocol-defined AEs to the Sponsor, investigators are required to promptly report to their respective IRB/EC all unanticipated problems involving risk to human patients. Some IRBs/ECs may want prompt notification of all SAEs, whereas others require notification only about events that are serious, assessed to be related to study treatment, and are unexpected. Investigators may receive written IND safety reports or other safety related communications from the Sponsor. Investigators are responsible for ensuring that such reports are reviewed and processed in accordance with regulatory requirements and with the policies and procedures established by their IRB/EC and archived in the site's study file.

#### 8.4 CONFIDENTIALITY

The Sponsor maintains confidentiality standards by coding each patient enrolled in the study through assignment of a unique patient identification number. This means that patient names are not included in data sets that are transmitted to any Sponsor location.

Patient medical information obtained by this study is confidential and may only be disclosed to third parties as permitted by the Informed Consent Form (or separate authorization for use and disclosure of personal health information) signed by the patient, unless permitted or required by law.

Medical information may be given to a patient's personal physician or other appropriate medical personnel responsible for the patient's welfare, for treatment purposes.

Data generated by this study must be available for inspection upon request by representatives of the U.S. FDA and other national and local health authorities, the Sponsor monitors, representatives, and collaborators, and the IRB/EC for each study site, as appropriate.

#### 8.5 FINANCIAL DISCLOSURE

Investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate health authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

# 9. <u>STUDY DOCUMENTATION, MONITORING, AND ADMINISTRATION</u>

#### 9.1 STUDY DOCUMENTATION

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented, including but not limited to the protocol, protocol amendments, Informed Consent Forms, and documentation of IRB/EC and governmental approval. In addition, at the end of the study, the investigator will receive the patient data, which includes an audit trail containing a complete record of all changes to data.

#### 9.2 SITE INSPECTIONS

Site visits will be conducted by the Sponsor or an authorized representative for inspection of study data, patients' medical records, and eCRFs. The investigator will permit national and local health authorities, the Sponsor monitors, representatives, and collaborators, and the IRBs/ECs to inspect facilities and records relevant to this study.

#### 9.3 ADMINISTRATIVE STRUCTURE

The study will have a SC, IDMC, central laboratory, IxRS, eCRF, and will be conducted by a contract research organization (CRO) together with the Sponsor.

### 9.4 PUBLICATION OF DATA AND PROTECTION OF TRADE SECRETS

The results of this study may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the Sponsor prior to submission. This allows the Sponsor to protect proprietary information and to provide comments based on information from other studies that may not yet be available to the investigator.

The Sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter trials only in their entirety and not as individual center data. In this case, a coordinating investigator will be designated by mutual agreement.

Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

Any formal publication of the study in which contribution the Sponsor personnel exceeded that of conventional monitoring will be considered as a joint publication by the investigator and the appropriate the Sponsor personnel.

Any inventions and resulting patents, improvements, and/or know-how originating from the use of data from this study will become and remain the exclusive and unburdened property of the Sponsor, except where agreed otherwise.

#### 9.5 PROTOCOL AMENDMENTS

Any protocol amendments will be prepared by the Sponsor. Protocol amendments will be submitted to the IRB/EC and to regulatory authorities in accordance with local regulatory requirements.

Approval must be obtained from the IRB/EC and regulatory authorities (as locally required) before implementation of any changes, except for changes necessary to eliminate an immediate hazard to patients or changes that involve logistical or administrative aspects only (e.g., change in Medical Monitor or contact information).

#### 10. REFERENCES

- International Agency for Research on Cancer. World Health Organization. GLOBOCAN 2012: Estimated cancer incidence, mortality and prevalence worldwide in 2012. <a href="http://globocan.iarc.fr/Pages/fact\_sheets\_cancer.aspx">http://globocan.iarc.fr/Pages/fact\_sheets\_cancer.aspx</a> (accessed 16 May 2014).
- 2. Sundaresan S, Penuel E, Sliwkowski MX. The biology of human epidermal growth factor receptor 2. Curr Oncol Rep 1999; 1:16–22.
- 3. Slamon DJ, Clark GM, Wong SG, et al. Human breast cancer; correlation of relapse and survival with amplification of the HER2/neo oncogene. Science 1987; 235:177–82.
- 4. Slamon DJ, Leyland-Jones B, Shak S, et al. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med 2001; 344:783–92.
- Marty M, Cognetti F, Maraninchi D, et al. Randomized Phase II trial of the efficacy and safety of trastuzumab combined with docetaxel in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer administered as first-line treatment: the M77001 study group. J Clin Oncol 2005; 23:4265–74.
- 6. Spector NL, Xia W, Burris H 3<sup>rd</sup>, et al. Study of the biologic effects of lapatinib, a reversible inhibitor of ErbB1 and ErbB2 tyrosine kinases, on tumor growth and survival pathways in patients with advanced malignancies. J Clin Oncol 2005; 23:2502–12.
- 7. Austin CD, De Mazière AM, Pisacane PI, et al. Endocytosis and sorting of ErbB2 and the site of action of cancer therapeutics trastuzumab and geldanamycin. Mol Biol Cell 2004; 15:5268–82.
- 8. Baselga J, Cortés J, et al; CLEOPATRA Study Group. Pertuzumab plus trastuzumab plus docetaxel for metastatic breast cancer. N Engl J Med 2012;366(2):109-19.
- 9. von Minckwitz G, du Bois A, Schmidt M, et al. Trastuzumab beyond progression in human epidermal growth factor receptor 2-positive advanced breast cancer: a german breast group 26/breast international group 03-05 study. J Clin Oncol 2009;27(12):1999-2006.
- Geyer CE, Forster J, Lindquist D, et al. Lapatinib plus capecitabine for HER2-positive advanced breast cancer. N Engl J Med 2006; 355:2733– 43.
- 11. Catalano V, Labianca R, Beretta GD, et al. Gastric cancer. Crit Rev Oncol Hematol 2005; 54:209–41.
- 12. Faivre J, Forman D, Esteve J, et al. Survival of patients with oesophageal and gastric cancers in Europe. Eur J Cancer 1998; 34:2167–75.
- 13. Power DG, Kelsen DP, Shah MA. Power Advanced gastric cancer--slow but steady progress. Cancer Treat Rev 2010; 36:384-92.
- 14. De Vivo R, Pignata S, Palaia R, et al. The role of chemotherapy in the management of gastric cancer. J Clin Gastroenterol 2000; 30:364–71.
- 15. Hofmann M, Stoss O, Shi D, et al. Assessment of a HER2 scoring system for gastric cancer: results from a validation study. Histopathology 2008; 52:797–805.
- Tanner M, Hollmen M, Junttila TT, et al. Amplification of HER2 in gastric cancer—association with topoisomerase IIa gene amplification, intestinal type, poor prognosis and sensitivity to trastuzumab. Ann Oncol 2005; 16:273–8.
- 17. Yoon HH, Shi Q, Sukov WR, et al. Association of HER2/ErbB2 expression and gene amplification with pathologic features and prognosis in esophageal adenocarcinomas. Clin Cancer Res 2012; 18:546–54.
- 18. Bang YJ, van Cutsem E, Feyereislova A, et al. Trastuzumab in combination with chemotherapy *versus* chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet 2010; 376:687–97.
- 19. Albarello L, Pecciarini L, Doglioni C. HER2 testing in gastric cancer. Adv Anat Pathol 2011; 18:53–9.
- 20. Junttila TT, Li G, Parsons K, et al. Trastuzumab-DM1 (T-DM1) retains all the mechanisms of action of trastuzumab and efficiently inhibits growth of lapatinib insensitive breast cancer. Breast Cancer Res Treat 2011; 128:347–56.
- 21. Issell BF, Crooke ST. Maytansine. Cancer Treat Rev 1978; 5:199-207.
- 22. Cassady JM, Chan KK, Floss HG, et al. Recent developments in the maytansinoid antitumor agents. Chem Pharm Bull (Tokyo) 2004; 52:1–26.
- 23. Cabanillas F, Chan KK, Floss HG, et al. Results of a Phase II study of maytansine in patients with breast carcinoma and melanoma. Cancer Treat Rep 1979; 63:507–9.
- 24. Erickson HK, Park PU, Widdison WC, et al. Antibody-maytansinoid conjugates are activated in targeted cancer cells by lysosomal degradation and linker-dependent intracellular processing. Cancer Res 2006; 66:4426–33.
- 25. Shen B-Q, Bumbaca D, Saad O, et al. Metabolic fate and pharmacokinetic characterization of trastuzumab emtansine (T-DM1): An emphasis on preclinical and clinical catabolism. ASCPT 2011.
- 26. Hurvitz SA, Dirix L, Kocsis J, et al. Phase II randomized study of trastuzumab emtansine versus trastuzumab plus docetaxel in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer. J Clin Oncol 2013;31(9):1157-63.
- 27. Verma S, Miles D, Gianni L, et al. Trastuzumab emtansine for HER2-positive advanced breast cancer. N Engl J Med 2012; 367:1783–91.

- 28. Krop IE, Kim SB, González-Martín A, et al. Trastuzumab emtansine versus treatment of physician's choice for pretreated HER2-positive advanced breast cancer (TH3RESA): a randomised, open-label, phase 3 trial. Lancet Oncol 2014;15(7):689-99.
- 29. Beeram M, Krop IE, Burris HA, et al. A phase 1 study of weekly dosing of trastuzumab emtansine (T-DM1) in patients with advanced human epidermal growth factor 2-positive breast cancer. Cancer 2012;118(23):5733-40.
- 30. Krop IE, Beeram M, Modi S, et al. Phase I study of trastuzumab-DM1, an HER2 antibody-drug conjugate, given every three weeks to patients with HER2-positive metastatic breast cancer. J. Clin Oncol 2010; 28:2698–704.
- 31. Burris HA 3rd, Rugo HS, Vukelja SJ, et al. Phase II study of the antibody drug conjugate trastuzumab-DM1 for the treatment of human epidermal growth factor receptor 2 (HER2)-positive breast cancer after prior HER2-directed therapy. J Clin Oncol 2011;29(4):398-405.
- 32. Krop IE, LoRusso P, Miller KD, et al. A phase II study of trastuzumab emtansine in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer who were previously treated with trastuzumab, lapatinib, an anthracycline, a taxane, and capecitabine. J Clin Oncol 2012;30(26):3234-41.
- 33. Gupta M, Wang B, Carrothers TJ, et al. Effects of trastuzumab emtansine (T-DM1) on QT interval and safety of pertuzumab plus T-DM1 in patients with previously treated human epidermal growth factor receptor 2-positive metastatic breast cancer. Clinical Pharm in Drug Dev 2013;2:11–24.
- 34. Therasse P, Eisenhauer EA, Verwij J. RECIST revisited: a review of validation studies on tumour assessment. Eur J Cancer 2000; 42:1031–9.
- 35. Gupta M, LoRusso PM, Wang B, et al. Clinical implications of pathophysiological and demographic covariates on the population pharmacokinetics of trastuzumab-DM1, a HER2-targeted antibody–drug conjugate, in patients with HER2-positive metastatic breast cancer. J Clin Pharmacol 2011; 52:691–703.
- 36. Girish S, Gupta M, Wang B, et al. Clinical pharmacology of trastuzumab emtansine (T-DM1): an antibody–drug conjugate in development for the treatment of HER2-positive cancer. Cancer Chemother Pharmacol 2012; 69:1229–40.
- 37. Igawa Y, Matsubara M, Matsunaga K, et al. Pharmacokinetic (PK) and pharmacodynamic (PD) analysis of trastuzumab emtansine (T-DM1) in Japanese patients with advanced or recurrent HER2-positive breast cancer (JO22591): Comparison with Western patients. ASCPT 2012.
- 38. Blum JL, Dieras V, Lo Russo PM, et al. Multicenter, Phase II study of oral capecitabine in taxane-pretreated metastatic breast carcinoma patients. Cancer 2001; 92:1759–68.

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 3, 30 June 2014

- 39. Blum JL, Jones SE, Buzdar AU, et al. Multicenter Phase II study of capecitabine in paclitaxel-refractory metastatic breast cancer. J Clin Oncol 1999; 17:485–93.
- 40. O'Shaughnessy J, Miles D, Vukelja S, Moiseyenko V, Ayoub JP, Cervantes G, Fumoleau P, Jones S, Lui WY, Mauriac L, Twelves C, Van Hazel G, Verma S, Leonard R. Superior survival with capecitabine plus docetaxel combination therapy in anthracycline-pretreated patients with advanced breast cancer: phase III trial results. J Clin Oncol 2002;20(12):2812-23.
- 41. Wardley A, Pivot X, Morales-Vasquez F, et al. Randomized phase II trial of first-line trastuzumab plus docetaxel and capecitabine compared with trastuzumab plus docetaxel in HER2-positive metastatic breast cancer. J Clin Oncol. 2010; 28:976-83.
- 42. Sawaki A, Ohashi Y, Omuro Y, et al. Efficacy of trastuzumab in Japanese patients with HER2-positive advanced gastric or gastroesophageal junction cancer: a subgroup analysis of the Trastuzumab for Gastric Cancer (ToGA) study. Gastric Cancer 2012; 15:313–22.
- 43. Lewis Phillips G, Fields CT, Crocker L, et al. Potent anti-tumor activity of trastuzumab-DM1 antibody conjugate in combination with cytotoxic chemotherapeutic agents, antibodies or small molecule kinase inhibitors. AACR 2008; poster#2133.
- 44. Press MF, Sauter G, Bernstein L, et al. Diagnostic evaluation of HER-2 as a molecular target: an assessment of accuracy and reproducibility of laboratory testing in large, prospective, randomized clinical trials. Clin Cancer Res 2005; 11:6598–607.
- 45. Gelmon KA, Vidal M, Sablin M-P, et al. Trastuzumab emtansine (T-DM1) plus capecitabine (X) in patients with HER2-positive MBC: MO28230 TRAX-HER2 phase 1 results. J Clin Oncol 32:5s, 2014 (suppl; abstr 606).
- 46. Yang J, Wang Y, Zhao H, et al. Combination of exposure-response and case-control analyses in regulatory decision making. J Clin Oncol 2011; 29: (Suppl); 4087.
- 47. Moldoveanu Z, Huang W-Q, Kulhavy R, et al. Human male genital tract secretions: both mucosal and systemic immune compartments contribute to the humoral immunity. J Immunol 2005; 175:4127–36.
- 48. Rubinstein LV, Korn EL, Freidlin B, et al. Design issues of randomized phase II trials and a proposal for phase II screening trials. J Clin Oncol 2005;23:7199–206.
- 49. Ratain MJ, Sargent DJ. Optimising the design of phase II oncology trials: the importance of radnomisation. Eur J Cancer 2009;45:275–80.

### Appendix 1 Schedule of Assessments

Table 1 Schedule of assessments for mBC patients (Phase I, Cohort 1 and Randomized Phase II)

| | Screening <sup>1</sup> | Cycle 1 | | Cycle 2–3 | | | Cycle 4 Onwards | | | Safety<br>Follow-Up<br>Visit | Follow-Up <sup>2</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 3-6<br>months |
| Informed Consent | Xª | | | | | | | | | | | |
| HER2 Status | Xp | | | | | | | | | | | |
| Medical History and Demographics | X | | | | | | | | | | | |
| Complete Physical Examination | X | | | | | | | | | | | |
| Limited Physical Examination <sup>c</sup> | | Х | | | Х | | | Х | | | Х | |
| Height and Weight <sup>d</sup> | X | Х | | | Х | | | Х | | | Х | |
| Vital Signs <sup>e</sup> | X | Х | | | Х | | | Х | | | Х | |
| ECOG Performance Status | Х | Х | | | Х | | | Х | | | Х | |
| Concomitant Medication Reporting | X <sup>f</sup> | Х | | | | | Ongoir | ng | | | | |
| AE Reporting | Xa | | | | | Ongoing | | | | | Х | X <sup>h</sup> |
| 12-lead ECG | X | | | | | | | | | | | |
| ECHO/MUGA <sup>i</sup> | Xi | | | Xi | | | Xi | | | Xi | Xi | |
| Tumor Assessments <sup>j</sup> | Х | | At Cycle 3 (9 weeks after randomization), and then every 4 <sup>th</sup> cycle (12 weeks thereafter, regardless of dose delay or early discontinuation) until PD or study termination, X whichever occurs earlier | | | | | | Х | | | |
| Brain CT or MRI <sup>k</sup> | Х | | | A | t the discre | etion of the | e investigat | tor, if clini | cally indica | ated, until I | PD | |
| Bone Scan/Imaging <sup>l</sup> | Х | | | | | | As clinicall | y indicate | d | | | |

Table 1 Schedule of assessments for mBC patients (Phase I, Cohort 1 and Randomized Phase II) (cont.)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | } | Cycl | e 4 Onwa | rds | Safety<br>Follow-Up<br>Visit | Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 3-6<br>months |
| Hematology <sup>m</sup> | Х | Xn | Xn | Xn | Xn | Xn | Xn | Xn | | | Х | |
| Biochemistryº | Х | Xn | Xn | Xn | Xn | Xn | Xn | Xn | | | Х | |
| Urinalysis <sup>p</sup> | Х | | As clinically indicated | | | | | | Х | | | |
| INR/aPTT | Х | F | As clinically indicated, e.g. for patients receiving anticoagulation therapy | | | | | | Х | | | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Χq | | | Χq | Х | Х |
| PK Samples (see <u>Appendix 2</u> ) <sup>r</sup> | | Xr | | | Xr | | | | | | | |
| Assessment of Patient<br>Hospitalizations and/or Hospital<br>Visits | | х | | | Х | | | Х | | | х | |
| Administration of Trastuzumab Emtansine | | D 2s | | | D 1s | | | D 1s | | | | |
| Administration of Capecitabine | | D 1 | 1–14 | | D 1 | _14 | | D 1 | _14 | | | |
| Overall Survival | | X | | | | | Х | Х | | | | |
| Randomization into the Phase II<br>Part of the Study | X <sup>t</sup> | | | | | | | | | | | |

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

- 1.NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within **14 days** prior to first treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1).
- 2.All patients will be followed-up every 6 months (except for pregnancy, which is at 3 and 6 months after safety follow-up visit until disease progresses for tumor assessment or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than PD will continue to undergo tumor assessments every 3–6 months.
- a)Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests.
- b)HER2-positivity is defined as IHC 3+ or gene amplification by ISH. It will be performed locally for patients with mBC.
- c)Limited symptom-directed physical examination.
- d)Height to be obtained at screening or at Cycle 1 Day 1 only.
- e)Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f)Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to first study treatment.
- g)During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h)Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatment-related AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i)Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, between Days 15 and 21 in cycles 1 and 3, and between Days 15 and 21 of every third cycle thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

- j)Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than PD, continued tumor assessments according to the protocol every 3–6 months until PD, withdrawal of consent, or study terminaton (whichever occurs earlier).
- k)Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 4 months) as detailed in Section 4.5.1.4 of the protocol and in Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- I)An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- m)Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and white blood cells (WBC) with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils.
- n)Assessments should be performed at screening, on Day 1, 8 and 15 of Cycles 1–3, on Day 1 of all subsequent cycles, and weekly following any hematologic AE. If capecitabine is discontinued due to toxicity, assessments should be performed weekly (minimum) until resolution of the AE (Grade ≤ 1/ baseline), and on Day 1 of subsequent cycles thereafter. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- o)Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, blood urea nitrogen (BUN)/urea (mandatory), creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN). p)Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.

- q)Serum β-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.
- r)Pharmacokinetic assessments will be performed during the MTD-Finding part of the study only (see Appendix 2).
- s)Trastuzumab emtansine will be administered on Day 1 of each 3-weekly cycle for all patients with mBC in Cohort 1 and Randomized Phase II period of the study except in the first cycle where trastuzumab emtansine will be given on Day 2 (to allow PK sampling).
- t)Patients will be randomized only in the Randomized Phase II part of the study. No blinding will be used, as this is an open-label study.

Table 2 Schedule of assessments for patients with LA/mGC (Phase I, Cohort 2)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | Cycle 4 Onwards | | | Safety<br>Follow-Up<br>Visit | Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28–42 days<br>after last<br>dose | every 3–6<br>months |
| Informed Consent | Xa | | | | | | | | | | | |
| HER2 Status | Xp | | | | | | | | | | | |
| Medical History and Demographics | Х | | | | | | | | | | | |
| Complete Physical Examination | Х | | | | | | | | | | | |
| Limited Physical Examination <sup>c</sup> | | Х | | | Х | | | Х | | | Х | |
| Height and Weight <sup>d</sup> | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | |
| Vital Signs <sup>e</sup> | Х | Х | | | Х | | | X | | | Х | |
| ECOG Performance Status | Х | Х | | | Х | | | Х | | | Х | |
| Concomitant Medication Reporting | X <sup>f</sup> | Х | | | | | Ongoi | ng | | | | |
| AE Reporting | Xa | | | | | Ongoing | | | | | Х | X <sup>h</sup> |
| 12-lead ECG | Х | | | | | | | | | | | |
| ECHO/MUGA <sup>i</sup> | Xi | | | Xi | | | Xi | | | Xi | Xi | |
| Tumor Assessments <sup>j</sup> | Х | At 9 we | At 9 weeks after C1D1, and every 12 weeks thereafter, regardless of dose delay or early discontinuation, until PD or study termination, whichever occurs earliest | | | | | | | | | |
| Brain CT or MRI <sup>k</sup> | Х | | | Α | t the disci | etion of the | e investiga | tor, if clinic | cally indica | ted, until F | סי | |
| Bone Scan/Imaging <sup>I</sup> | Х | | | | | | As clinical | ly indicate | d | | | |

| Hematology <sup>m</sup> | Χ | Xn | Xn | Xn | Xn | Xn | Xn | Xn | Xn | X <sup>n</sup> | Χ | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Biochemistry <sup>o</sup> | Х | Xn | Xn | Xn | Xn | Xn | X <sup>n</sup> | Xn | Xn | X <sup>n</sup> | Х | |
| Urinalysis <sup>p</sup> | Х | | • | • | As c | inically ind | dicated | • | | | Х | |
| INR/aPTT | Х | А | s clinicall | y indicate | d, e.g. for | patients r | eceiving an | ticoagulat | ion therap | у | Х | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Χq | | | Χq | Х | Х |
| PK/PD Samples (see Appendix 2) | | Х | | | Х | | | | | | | |
| Assessment of Patient Hospitalizations and/or Hospital Visits | | Х | | | х | | | Х | | | Х | |
| Administration of Trastuzumab<br>Emtansine | | D 2 <sup>r</sup> | х | х | х | Х | х | Х | Х | Х | | |
| Administration of Capecitabine | | D 1- | -14 | | D 1 | -14 | | D 1 | -14 | | | |
| Overall Survival | | X | | | | | Х | Х | | | | |

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

- 1.NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within **14 days** prior to first study treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1) visit.
- 2.All patients will be followed-up every 6 months (except for pregnancy, which is at 3 and 6 months after safety follow-up visit) until disease progresses for tumor assessment or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than PD will continue to undergo tumor assessments every 3–6 months.
- a)Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests.
- b)HER2-positivity is defined as IHC 3+ alone or IHC 2+ in combination with gene amplification by ISH. For patients with mGC enrolled into Cohort 2, central confirmation of HER2 status is required.
- c)Limited symptom-directed physical examination.
- d)Height to be obtained at screening or at Cycle 1 Day 1 only.
- e)Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f)Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to fist study treatment.
- g)During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h)Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatment-related AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i)Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, between Days 15 and 21 in cycles 1 and 3, and between Days 15 and 21 of every 3rd cycle thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

# Study MO28230

- j)Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than PD, continue tumor assessments according to the protocol every 3–6 months until PD, withdrawal of consent, or study termination (whichever occurs earliest).
- k)Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 4 months) as detailed in Section 4.5.1.4 of the protocol and in Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- I)An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to first study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- m)Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and WBC with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils).
- n)Assessments should be performed at screening, on Day 1, 8 and 15 of all cycles. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- o)Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, BUN/urea (mandatory), creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN).
- p)Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.
- q)Serum β-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.
- r)Trastuzumab emtansine will be administered on Day 1 of each weekly cycle for all patients enrolled in Cohort 2 (A&B) except in the first cycle where trastuzumab emtansine will be given on DAY 2 (to allow drug interaction assessment).

# Appendix 2 Pharmacokinetic Sampling for Phase I, Metastatic Breast and Gastric Cancer Patients

| | Trastuzumab<br>emtansine, total<br>trastuzumab and DM1ª<br>PK samples (serum) | Capecitabine and 5-FU<br>PK samples (plasma) |
|---|---|---|
| Cycle 1 Day 1 | | |
| Pre-capecitabine dose | | Х |
| 30 min post capecitabine dosing | | X |
| 60 min post capecitabine dosing | | X |
| 1.5 hours post capecitabine dosing | | х |
| 2 hours post capecitabine dosing | | x |
| 2.5 hours post capecitabine dosing | | x |
| 4 hours post capecitabine dosing | | x |
| 6 hours post capecitabine dosing | | х |
| Cycle 1 Day 2 | | |
| Pre-trastuzumab emtansine dose | х | |
| 15-30 min after end of trastuzumab emtansine infusion | х | |
| Pre-capecitabine dose | | X |
| 30 min post capecitabine dosing | | X |
| 2 hours post capecitabine dosing | | х |
| 6 hours post capecitabine dosing | | x |
| Cycle 1 Day 3 | | |
| 24 hours (± 2 hours) after the end of infusion of trastuzumab emtansine | х | |
| Cycle 1 Day 9 | | |
| 7 days (± 1 day) after the end of infusion of trastuzumab emtansine <sup>a</sup> | х | |
| Cycle 2 Day 1 | | |
| Pre- capecitabine and trastuzumab emtansine dose <sup>a</sup> | x | |
| 15–30 min after end of trastuzumab emtansine infusion | х | |

### Trastuzumab emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 3, 30 June 2014

| | х |
|---|---|
| | Х |
| | х |
| | х |
| | х |
| | х |
| | х |
| х | |
| x | |
| × | |
| | x |

PK = pharmacokinetic; 5-FU = 5-fluoruracil

Data from historic studies have determined that results are the lower limit of quantitation.

<sup>&</sup>lt;sup>a</sup> = Plasma DM1 samples will not be collected at Day 7 post-infusion of trastuzumab emtansine neither at pre-dose of Cycle 2 and Cycle 3.

Selected sections from the Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1,<sup>1</sup> are presented below, with slight modifications and the addition of explanatory text as needed for clarity.<sup>2</sup>

### Measurability of Tumor at Baseline

#### **Definitions**

At baseline, tumor lesions/lymph nodes will be categorized as measurable or non-measurable as described below.

#### a. Measurable Tumor Lesions

**Tumor Lesions.** Tumor lesions must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size as follows:

- 10 mm by CT or magnetic resonance imaging (MRI) scan (CT/MRI scan slice thickness/interval no greater than 5 mm)
- 10mm caliper measurement by clinical examination (lesions that cannot be accurately measured with calipers should be recorded as nonmeasurable)
- 20 mm by chest X-ray

**Malignant Lymph Nodes.** To be considered pathologically enlarged and measurable, a lymph node must be  $\geq$  15 mm in the short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and follow-up, only the short axis will be measured and followed. See also notes below on "Baseline Documentation of Target and Non-Target Lesions" for information on lymph node measurement.

<sup>&</sup>lt;sup>1</sup> Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (Version 1.1). Eur J Cancer 2009;45:228–47.

<sup>&</sup>lt;sup>2</sup> For consistency within this document, the section numbers and cross-references to other sections within the article have been deleted and minor formatting changes have been made.

#### b. Non-Measurable Tumor Lesions

Non-measurable tumor lesions encompass small lesions (longest diameter > 10 mm or pathological lymph nodes with short axis ≥ 10 but < 15 mm) as well as truly non-measurable lesions. Lesions considered truly non-measurable include leptomeningeal disease, ascites, pleural or pericardial effusion, inflammatory breast disease, lymphangitic involvement of skin or lung, peritoneal spread, and abdominal mass/abdominal organomegaly identified by physical examination that is not measurable by reproducible imaging techniques.

### c. Special Considerations Regarding Lesion Measurability

Bone lesions, cystic lesions, and lesions previously treated with local therapy require particular comment, as outlined below.

#### Bone Lesions:

- Bone scan, PET scan, or plain films are not considered adequate imaging techniques for measuring bone lesions. However, these techniques can be used to confirm the presence or disappearance of bone lesions.
- Lytic bone lesions or mixed lytic-blastic lesions, with identifiable soft tissue components, that can be evaluated by cross-sectional imaging techniques such as CT or MRI can be considered as measurable lesions if the soft tissue component meets the definition of measurability described above.
- Blastic bone lesions are non-measurable.

### Cystic Lesions:

- Lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor non-measurable) since they are, by definition, simple cysts.
- Cystic lesions thought to represent cystic metastases can be considered
  as measurable lesions, if they meet the definition of measurability
  described above. However, if non-cystic lesions are present in the same
  patient, these are preferred for selection as target lesions.

#### Lesions with Prior Local Treatment:

 Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion. Study protocols should detail the conditions under which such lesions would be considered measurable.

### **Target Lesions: Specifications by Methods of Measurements**

#### a. Measurement of Lesions

All measurements should be recorded in metric notation, using calipers if clinically assessed. All baseline evaluations should be performed as close as possible to the treatment start and never more than 28 days before the beginning of the treatment.

#### b. Method of Assessment

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during the study. Imaging-based evaluation should always be the preferred option.

**Clinical Lesions.** Clinical lesions will only be considered measurable when they are superficial and ≥ 10 mm in diameter as assessed using calipers (e.g., skin nodules). For the case of skin lesions, documentation by color photography including a ruler to estimate the size of the lesion is suggested.

**Chest X-Ray.** Chest CT is preferred over chest X-ray, particularly when progression is an important endpoint, since CT is more sensitive than X-ray, particularly in identifying new lesions. However, lesions on chest X-ray may be considered measurable if they are clearly defined and surrounded by aerated lung.

**CT, MRI.** CT is the best currently available and reproducible method to measure lesions selected for response assessment. This guideline has defined measurability of lesions on CT scan based on the assumption that CT slice thickness is 5 mm or less. When CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness. MRI is also acceptable.

If prior to enrollment it is known that a patient is unable to undergo CT scans with IV contrast because of allergy or renal insufficiency, the decision as to whether a non-contrast CT or MRI (without IV contrast) will be used to evaluate the patient at baseline and during the study should be guided by the tumor type under investigation and the anatomic location of the disease. For patients who develop contraindications to contrast after baseline contrast CT is done, the decision as to whether non-contrast CT or MRI (enhanced or non-enhanced) will be performed should also be based on the tumor type and the anatomic location of the disease, and should be optimized to allow for comparison with the prior studies if possible. Each case should be discussed with the radiologist to determine if substitution of these other approaches is possible and, if not, the patient should be considered not evaluable from that point forward. Care must

be taken in measurement of target lesions on a different modality and interpretation of non-target disease or new lesions, since the same lesion may appear to have a different size using a new modality.

**Ultrasound.** Ultrasound is not useful in assessment of lesion size and should not be used as a method of measurement.

**Endoscopy, Laparoscopy, Tumor Markers, Cytology, Histology.** The utilization of these techniques for objective tumor evaluation cannot generally be advised.

### **Tumor Response Evaluation**

#### Assessment of Overall Tumor Burden and Measurable Disease

To assess objective response or future progression, it is necessary to estimate the overall tumor burden at baseline and use this as a comparator for subsequent measurements. Measurable disease is defined by the presence of at least one measurable lesion, as detailed above.

### **Baseline Documentation of Target and Non-Target Lesions**

When more than one measurable lesion is present at baseline, all lesions up to a maximum of five lesions total (and a maximum of two lesions per organ) representative of all involved organs should be identified as target lesions and will be recorded and measured at baseline. This means that, for instances in which patients have only one or two organ sites involved, a maximum of two lesions (one site) and four lesions (two sites), respectively, will be recorded. Other lesions (albeit measurable) in those organs will be recorded as non-measurable lesions (even if the size is > 10 mm by CT scan).

Target lesions should be selected on the basis of their size (lesions with the longest diameter) and be representative of all involved organs, but in addition should lend themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion does not lend itself to reproducible measurement, in which circumstance the next largest lesion that can be measured reproducibly should be selected.

Lymph nodes merit special mention since they are normal anatomical structures that may be visible by imaging even if not involved by tumor. As noted above, pathological nodes that are defined as measurable and may be identified as target lesions must meet the criterion of a short axis of  $\geq 15$  mm by CT scan. Only the short axis of these nodes will contribute to the baseline sum. The short axis of the node is the diameter normally used by radiologists

to judge if a node is involved by solid tumor. Nodal size is normally reported as two dimensions in the plane in which the image is obtained (for CT this is almost always the axial plane; for MRI the plane of acquisition may be axial, sagittal, or coronal). The smaller of these measures is the short axis. For example, an abdominal node that is reported as being 20 mm × 30 mm has a short axis of 20 mm and qualifies as a malignant, measurable node. In this example, 20 mm should be recorded as the node measurement. All other pathological nodes (those with short axis ≥ 10 mm but < 15 mm) should be considered non-target lesions. Nodes that have a short axis of < 10 mm are considered non-pathological and should not be recorded or followed.

A sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the baseline sum of diameters. If lymph nodes are to be included in the sum, then, as noted above, only the short axis is added into the sum. The baseline sum of diameters will be used as a reference to further characterize any objective tumor regression in the measurable dimension of the disease.

All other lesions (or sites of disease), including pathological lymph nodes, should be identified as non-target lesions and should also be recorded at baseline. Measurements are not required and these lesions should be followed as "present," "absent," or in rare cases "unequivocal progression."

In addition, it is possible to record multiple non-target lesions involving the same organ as a single item on the Case Report Form (CRF) (e.g., "multiple enlarged pelvic lymph nodes" or "multiple liver metastases").

### **Response Criteria**

### a. Evaluation of Target Lesions

This section provides the definitions of the criteria used to determine objective tumor response for target lesions.

- Complete response (CR): Disappearance of all target lesions
   Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.</li>
- Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters
- Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline

In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.

The appearance of one or more new lesions is also considered progression.

 Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study

### b. Special Notes on the Assessment of Target Lesions

**Lymph Nodes.** Lymph nodes identified as target lesions should always have the actual short axis measurement recorded (measured in the same anatomical plane as the baseline examination), even if the nodes regress to < 10 mm on study. This means that when lymph nodes are included as target lesions, the sum of lesions may not be zero even if CR criteria are met, since a normal lymph node is defined as having a short axis of < 10 mm.

Target Lesions That Become Too Small to Measure. During the study, all lesions (nodal and non-nodal) recorded at baseline should have their actual measurements recorded at each subsequent evaluation, even when very small (e.g., 2 mm). However, sometimes lesions or lymph nodes that are recorded as target lesions at baseline become so faint on CT scan that the radiologist may not feel comfortable assigning an exact measure and may report them as being too small to measure. When this occurs, it is important that a value be recorded on the CRF, as follows:

- If it is the opinion of the radiologist that the lesion has likely disappeared, the measurement should be recorded as 0 mm.
- If the lesion is believed to be present and is faintly seen but too small to measure, a default value of 5 mm should be assigned and below measurable limit (BML) should be ticked. (Note: It is less likely that this rule will be used for lymph nodes since they usually have a definable size when normal and are frequently surrounded by fat such as in the retroperitoneum; however, if a lymph node is believed to be present and is faintly seen but too small to measure, a default value of 5 mm should be assigned in this circumstance as well and BML should also be ticked).

To reiterate, however, if the radiologist is able to provide an actual measure, that should be recorded, even if it is below 5 mm, and in that case BML should not be ticked.

**Lesions That Split or Coalesce on Treatment.** When non-nodal lesions fragment, the longest diameters of the fragmented portions should be added

together to calculate the target lesion sum. Similarly, as lesions coalesce, a plane between them may be maintained that would aid in obtaining maximal diameter measurements of each individual lesion. If the lesions have truly coalesced such that they are no longer separable, the vector of the longest diameter in this instance should be the maximum longest diameter for the coalesced lesion.

### c. Evaluation of Non-Target Lesions

This section provides the definitions of the criteria used to determine the tumor response for the group of non-target lesions. While some non-target lesions may actually be measurable, they need not be measured and instead should be assessed only qualitatively at the time points specified in the protocol.

- Complete response (CR): Disappearance of all non-target lesions and (if applicable) normalization of tumor marker level
  - All lymph nodes must be non-pathological in size (< 10 mm short axis).
- Non-CR/Non-PD: Persistence of one or more non-target lesions and/or (if applicable) maintenance of tumor marker level above the normal limits
- Progressive disease (PD): Unequivocal progression of existing non-target lesions

The appearance of one or more new lesions is also considered progression.

### d. Special Notes on Assessment of Progression of Non-Target Disease

When the Patient Also Has Measurable Disease. In this setting, to achieve unequivocal progression on the basis of the non-target disease, there must be an overall level of substantial worsening in non-target disease in a magnitude that, even in the presence of SD or PR in target disease, the overall tumor burden has increased sufficiently to merit discontinuation of therapy. A modest increase in the size of one or more non-target lesions is usually not sufficient to qualify for unequivocal progression status. The designation of overall progression solely on the basis of change in non-target disease in the face of SD or PR of target disease will therefore be extremely rare.

When the Patient Has Only Non-Measurable Disease. This circumstance arises in some Phase III trials when it is not a criterion of study entry to have measurable disease. The same general concepts apply here as noted above; however, in this instance there is no measurable disease assessment to factor into the interpretation of an increase in non-measurable disease burden. Because worsening in non-target disease cannot be easily quantified (by definition: if all lesions are truly non-measurable), a useful test that can be

applied when assessing patients for unequivocal progression is to consider if the increase in overall disease burden based on the change in non-measurable disease is comparable in magnitude to the increase that would be required to declare PD for measurable disease, that is, an increase in tumor burden representing an additional 73% increase in volume (which is equivalent to a 20% increase in diameter in a measurable lesion). Examples include an increase in a pleural effusion from "trace" to "large" or an increase in lymphangitic disease from localized to widespread, or may be described in protocols as "sufficient to require a change in therapy." If unequivocal progression is seen, the patient should be considered to have had overall PD at that point. While it would be ideal to have objective criteria to apply to non-measurable disease, the very nature of that disease makes it impossible to do so; therefore, the increase must be substantial.

#### e. New Lesions

The appearance of new malignant lesions denotes PD; therefore, some comments on detection of new lesions are important. There are no specific criteria for the identification of new radiographic lesions; however, the finding of a new lesion should be unequivocal, that is, not attributable to differences in scanning technique, change in imaging modality, or findings thought to represent something other than tumor (e.g., some "new" bone lesions may be simply healing or flare of pre-existing lesions). This is particularly important when the patient's baseline lesions show partial or CR. For example, necrosis of a liver lesion may be reported on a CT scan report as a "new" cystic lesion, which it is not.

A lesion identified during the study in an anatomical location that was not scanned at baseline is considered a new lesion and will indicate PD.

If a new lesion is equivocal, e.g., because of its small size, continued therapy and follow-up evaluation will clarify if it represents truly new disease. If repeat scans confirm there is definitely a new lesion, then progression should be declared using the date of the initial scan.

#### **Evaluation of Response**

### a. Time Point Response (Overall Response)

It is assumed that at each protocol-specified time point, a response assessment occurs. **Table 1** provides a summary of the overall response status calculation at each time point for patients who have measurable disease at baseline.

When patients have non-measurable (therefore non-target) disease only, **Table 2** is to be used.

Table 1 Time Point Response: Patients with Target Lesions (with or without Non-Target Lesions)

| Target Lesions | Non-Target Lesions | New Lesions | Overall Response |
|---|---|---|---|
| | CR | No | CR |
| CR | | | |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | NE |
| PD | Any | Yes or no | PD |
| Any | PD | Yes or no | PD |
| Any | Any | Yes | PD |

$$\label{eq:crossing} \begin{split} &\text{CR=complete response; NE=not evaluable; PD=progressive disease; PR=partial response; SD=stable disease.} \end{split}$$

Table 2 Time Point Response: Patients with Non-Target Lesions Only

| Non-Target Lesions | New Lesions | Overall Response |
|--------------------|-------------|------------------|
| | No | CR |
| CR | | |
| Non-CR/non-PD | No | Non-CR/non-PD a |
| Not all evaluated | No | NE |
| Unequivocal PD | Yes or no | PD |
| Any | Yes | PD |

CR=complete response; NE=not evaluable; PD=progressive disease.

a "Non-CR/non-PD" is preferred over "stable disease" for non-target disease since stable disease is increasingly used as an endpoint for assessment of efficacy in some trials; thus, assigning "stable disease" when no lesions can be measured is not advised.

### b. Missing Assessments and Not Evaluable Designation

When no imaging/measurement is done at all at a particular time point, the patient is not evaluable at that time point. If only a subset of lesion measurements are made at an assessment, usually the case is also considered not evaluable at that time point, unless a convincing argument can be made that the contribution of the individual missing lesion(s) would not change the assigned time point response. This would be most likely to happen in the case of PD. For example, if a patient had a baseline sum of 50 mm with three measured lesions and during the study only two lesions were assessed, but those gave a sum of 80 mm, the patient will have achieved PD status, regardless of the contribution of the missing lesion.

If one or more target lesions were not assessed either because the scan was not done or the scan could not be assessed because of poor image quality or obstructed view, the response for target lesions should be "unable to assess" since the patient is not evaluable. Similarly, if one or more non-target lesions are not assessed, the response for non-target lesions should be "unable to assess" except where there is clear progression. Overall response would be "unable to assess" if either the target response or the non-target response is "unable to assess" except where this is clear evidence of progression, as this equates with the case being not evaluable at that time point.

#### c. Special Notes on Response Assessment

When nodal disease is included in the sum of target lesions and the nodes decrease to "normal" size (<10 mm), they may still have a measurement reported on scans. This measurement should be recorded even though the nodes are normal in order not to overstate progression should it be based on increase in size of the nodes. As noted earlier, this means that patients with CR may not have a total sum of "zero" on the CRF.

Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of PD at that time should be reported as "symptomatic deterioration." Every effort should be made to document objective progression even after discontinuation of treatment. Symptomatic deterioration is not a descriptor of an objective response; it is a reason for stopping study therapy. The objective response status of such patients is to be determined by evaluation of target and non-target disease as shown in **Table 1**, **Table 2**, **Table 3**.

Table 3 Best Overall Response When Confirmation Is Required

| Overall Response at First Time Point | Overall Response at<br>Subsequent Time Point | Best Overall Response |
|---|---|---|
| Time Femi | CR | CR |
| CR | OI C | OIC |
| CR | PR | SD, PD, or PR <sup>a</sup> |
| CR | SD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| CR | PD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| CR | NE | SD, provided minimum<br>duration for SD was met;<br>otherwise, NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| PR | NE | SD, provided minimum<br>duration for SD was met;<br>otherwise, NE |
| NE | NE | NE |

CR=complete response; NE=not evaluable; PD=progressive disease; PR=partial response; SD=stable disease.

a If a CR is truly met at the first time point, any disease seen at a subsequent time point, even disease meeting PR criteria relative to baseline, qualifies as PD at that point (since disease must have reappeared after CR). Best response would depend on whether the minimum duration for SD was met. However, sometimes CR may be claimed when subsequent scans suggest small lesions were likely still present and in fact the patient had PR, not CR, at the first time point. Under these circumstances, the original CR should be changed to PR and the best response is PR.

For equivocal findings of progression (e.g., very small and uncertain new lesions; cystic changes or necrosis in existing lesions), treatment may continue until the next scheduled assessment. If at the next scheduled assessment, progression is confirmed, the date of progression should be the earlier date when progression was suspected.

In studies for which patients with advanced disease are eligible (i.e., primary disease still or partially present), the primary tumor should also be captured as a target or non-target lesion, as appropriate. This is to avoid an incorrect assessment of CR if the primary tumor is still present but not evaluated as a target or non-target lesion.

### Appendix 4 Instructions for Scans in the Event of Isotope Shortage

Two key suppliers of Tc-99m generators (Chalk River Reactor, Canada and High Flux Reactor, the Netherlands) are expected to close. Supplies from other reactor sources will be unable to meet the expected world-wide patient-care needs. As a result, significant shortages of Tc-99m are expected, and the instructions listed below should be followed:

- ECHO will be the preferred imaging modality over MUGA scans to evaluate cardiac function.
- Tc-99m bone scans should be obtained as part of the baseline tumor assessment in all patients and should be repeated to confirm a CR or if progression of existing bone lesions and/or the development of new bone lesions is clinically suspected.
  - If a bone scan cannot be performed at baseline or if the investigator suspects that a bone scan may not be able to be repeated during the course of the study because of the Tc-99m shortage, the investigator may choose F-18 NaF or FDG-PET scan as an alternative.
- If bone lesions are selected as index non-target lesions, they must be apparent on baseline CT scans or other radiographic modalities (e.g., skeletal X-rays that can be repeated in subsequent tumor assessments). Additional scans may be obtained to follow clinically important bone lesions if not visualized on the chest, abdomen, or pelvic CT scan.

These measures are intended to ensure that the same method of assessment and the same imaging technique is used throughout the study for each patient. If there is a question regarding the choice of alternatives in the event that a standard bone scan cannot be obtained during screening and/or during the study, please contact the Medical Monitor.

# Appendix 5 New York Heart Association Classification of Functional Cardiac Capacity

| Class | |
|---|---|
| I | No limitation: Ordinary physical activity does not cause undue fatigue, dyspnea, or palpitation. |
| II | Slight limitation of physical activity: Such patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitations, dyspnea, or angina. |
| III | Marked limitation of physical activity: Although patients are comfortable at rest, less than ordinary physical activity will lead to symptoms. |
| IV | Inability to carry on physical activity without discomfort: Symptoms of congestive heart failure are present even at rest. With any physical activity, increased discomfort is experienced. |

From: Criteria Committee, New York Heart Association, Inc. Diseases of the heart and blood vessels. Nomenclature and criteria for diagnosis. 6th ed. Boston, Little, Brown and Co, 1964:114.

### Appendix 6 ECOG Performance Status

| | Scale |
|---|---|
| Grade | |
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, i.e., light housework, office work |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair |
| 5 | Dead |

50. http://www.ecog.org/general/perf\_stat.html

#### PROTOCOL

TITLE: PHASE I STUDY OF THE COMBINATION OF TRASTUZUMAB EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED/METASTATIC GASTRIC CANCER PATIENTS, FOLLOWED BY A RANDOMIZED, OPEN-LABEL PHASE II STUDY OF TRASTUZUMAB EMTANSINE AND CAPECITABINE VERSUS TRASTUZUMAB EMTANSINE ALONE IN HER2-POSITIVE

PROTOCOL NUMBER: MO28230 VERSION NUMBER: 4

**EUDRACT NUMBER:** 2012-001547-46


Capecitabine (RO091978)

MEDICAL MONITOR: MD

SPONSOR: F. Hoffmann-La Roche Ltd

**METASTATIC BREAST CANCER** 

DATE FINAL: Last date of signatures below

#### FINAL PROTOCOL APPROVAL

Name
Date and signature

22.3. 16

Statistician

23 Marcl 2016


The information contained in this document, especially any unpublished data, is the property of F. Hoffmann-La Roche Ltd (or under its control) and therefore is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Ethics Committee or Institutional Review Board. It is understood that this information will not be disclosed to others without written authorization from Roche except to the extent necessary to obtain informed consent from persons to whom the drug may be administered.

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 4, 23 Mar 2016

### **TABLE OF CONTENTS**

| PR | OTOCOL ACC | CEPTANCE FORM | 10 |
|---|---|---|---|
| PRO | OTOCOL SYN | IOPSIS | 11 |
| 1. | BACKGROU | ND | 28 |
| | 1.1 | Background on Disease | 28 |
| | 1.1.1 | HER2-Positive Breast Cancer | 28 |
| | 1.1.2<br>Gastric Ca | HER2-Positive Locally Advanced/Metastatic ncer | 29 |
| | 1.2 | Background on Study Drugs | 30 |
| | 1.2.1 | Trastuzumab Emtansine | 30 |
| | 1.2.1.1 | Study TDM3569g | 32 |
| | 1.2.1.2 | Study TDM4258g | 32 |
| | 1.2.1.3 | Study TDM4374g | 33 |
| | 1.2.1.4 | Study TDM4450g | 34 |
| | 1.2.1.5 | Study TDM4688g | 35 |
| | 1.2.1.6 | Phase III Study TDM4370g | 35 |
| | 1.2.1.7 | Phase III study TDM4997g | 36 |
| | 1.2.1.8 | Pharmacokinetics | 37 |
| | 1.2.2 | Capecitabine | 38 |
| | 1.2.2.1<br>Trastuz | Study BO18255: Capecitabine and rumab in LA/mGC | 39 |
| | 1.2.3<br>Trastuzum | Preclinical Data of the Combination of ab Emtansine and a Fluoropyrimidine | 40 |
| | 1.3 | Study Rationale and Risk-Benefit Assessment | 42 |
| | 1.3.1 | For mBC | 42 |
| | 1.3.2 | For mGC | 43 |
| 2. | OBJECTIVE | S | 44 |
| | 2.1 | Phase I: MTD-Finding of Trastuzumab Emtansine and Capecitabine in mBC | 44 |
| | 2.1.1 | Primary Objective | 44 |
| | 2.1.2 | Secondary Objectives | 44 |
| | 2.2 | Randomized Phase II: Exploration of Efficacy and Safety in mBC | 11 |
| | 2.2.1 | Primary Objective | |
| | 2.2.2 | Secondary Objectives | |
| | tuzumab Emtar | nsine—F. Hoffmann-La Roche Ltd<br>/ersion 4, 23 Mar 2016 | 2 |

3

| 020 | | | Study MO28230 |
|---|---|---|---|
| | 2.3 | Phase I: MTD Finding of Trastuzumab<br>Emtansine and Capecitabine in LA/mGC | 45 |
| | 2.3.1 | Primary Objective | 45 |
| | 2.3.2 | Secondary Objectives | |
| 3. | STUDY DES | IGN | 45 |
| 0. | 3.1 | Description of Study | |
| | 3.1.1 | Overview of Study Design | |
| | 3.1.1.1<br>mBC | | |
| | | Overview of Phase II: Exploration of Efficacy fety in Patients with mBC | |
| | 3.1.1.3<br>Patients | Overview of Phase I Design in LA/mGC s 50 | |
| | 3.1.1.4 | Number of Patients | 51 |
| | 3.1.1.5 | Number of Centers | 51 |
| | 3.1.2 | Steering Committee | 51 |
| | 3.1.3 | Independent Data Monitoring Committee | 51 |
| | 3.2 | End of Study | 51 |
| | 3.3 | Rationale for Study Design | 52 |
| | 3.3.1 | Rationale for Patient Group Selection | 52 |
| | 3.3.1.1 | Rationale for Phase I | 52 |
| | 3.3.1.2 | Rationale for Randomized Phase II | 53 |
| | 3.3.2<br>Selection | Rationale for Investigational Medicinal Dose 53 | |
| | 3.3.2.1 | In Patients with mBC | 53 |
| | 3.3.2.2 | In Patients with mGC | 53 |
| | 3.3.2.3 | Rationale for Duration of Treatment | 54 |
| | 3.3.3 | Pharmacokinetic Sampling Rationale | 54 |
| | 3.4 | Outcome Measures | 55 |
| | 3.4.1 | Phase I: mBC | 55 |
| | 3.4.1.1 | Primary Outcome Measure | 55 |
| | 3.4.1.2 | Secondary Outcome Measure | 55 |
| | 3.4.1.3 | Primary Safety Outcome Measure | 55 |
| | 3.4.1.4 | Secondary Safety Outcome Measures | 55 |
| | 3.4.1.5 | Pharmacokinetic Outcome Measures | 55 |

Kadcyla (RO5304020) Roche Clinical Study Report - Protocol MO28230 Research Report 1078906 1563

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 4, 23 Mar 2016

Randomized Phase II: Exploration of Efficacy

and Safety in mBC......56

| | 3.4.2.1 | Primary Efficacy Outcome Measure | 56 |
|---|---|---|---|
| | 3.4.2.2 | Secondary Efficacy Outcome Measures | 56 |
| | 3.4.2.3 | Primary Safety Outcome Measure | 56 |
| | 3.4.2.4 | Secondary Safety Outcome Measures | 56 |
| | 3.4.2.5 | Pharmacokinetic Outcome Measures | . 57 |
| | 3.4.3 | Phase I: LA/mGC | . 57 |
| | 3.4.3.1 | Primary Outcome Measure | . 57 |
| | 3.4.3.2 | Secondary Efficacy Outcome Measure | . 57 |
| | 3.4.3.3 | Secondary Safety Outcome Measures | . 57 |
| | 3.4.3.4 | Pharmacokinetic Outcome Measures | . 58 |
| 4. | MATERIALS | AND METHODS | . 58 |
| | 4.1 | Patients | . 58 |
| | 4.1.1 | Patients with mBC | . 58 |
| | 4.1.2 | LA/mGC Patients | . 58 |
| | 4.1.3 | Inclusion Criteria | . 59 |
| | 4.1.3.1 | For Patients with mBC | . 59 |
| | 4.1.3.2 | For Patients with LA/mGC | 60 |
| | 4.1.4 | Exclusion Criteria | 62 |
| | 4.1.4.1 | For Patients with mBC | 62 |
| | 4.1.4.2 | For Patients with LA/mGC | 63 |
| | 4.1.5 | Patient Replacement Policy | 65 |
| | 4.2 | Method of Treatment Assignment | 65 |
| | 4.3 | Study Treatment | 65 |
| | 4.3.1 | Formulation, Packaging, and Handling | 65 |
| | 4.3.1.1 | Trastuzumab Emtansine | 65 |
| | 4.3.1.2 | Capecitabine | 66 |
| | 4.3.2 | Dosage and Administration | 67 |
| | | For Patients with mBC | |
| | 4.3.2.2 | For Patients with LA/mGC | . 68 |
| | 4.3.3 | Investigational Medicinal Product | 60 |
| | 4.3.4 | ility Post-trial Access to Extension Study | |
| | 4.3.4 | Concomitant And Excluded Therapies | |
| | 4.4.1 | Permitted Therapy | |
| | 4.4.1 | Prohibited Therapy | 69 |
| | <b></b> / | TO THE PROPERTY OF THE PROPERT | 1151 |

| | 4.5 | Study Assessments | 70 |
|---|---|---|---|
| | 4.5.1 | Description of Study Assessments | 70 |
| | 4.5.1.1 | Medical History and Demographic Data | 70 |
| | 4.5.1.2 | Vital Signs | 71 |
| | 4.5.1.3 | Physical Examinations | 71 |
| | 4.5.1.4 | Tumor and Response Evaluations | 71 |
| | 4.5.1.5 | Laboratory Assessments | 72 |
| | 4.5.1.6 | Electrocardiograms | 73 |
| | 4.5.1.7 | ECOG Performance Status | 73 |
| | 4.5.1.8 | ECHO/MUGA | 73 |
| | 4.5.2 | Timing of Study Assessments | 73 |
| | 4.5.2.1 | Screening and Pretreatment Assessments | 73 |
| | 4.5.2.2 | Assessments during Treatment | 74 |
| | 4.5.2.3<br>Termina | Assessments at Study Completion/Early ation Visit | 75 |
| | 4.5.2.4 | Follow-up Assessments | 75 |
| | 4.5.2.5 | Assessments at Unplanned Visits | 75 |
| | 4.6 | Patient and STUDY Discontinuation | 75 |
| | 4.6.1 | Patient Discontinuation | 75 |
| | 4.6.2 | Study Discontinuation | 76 |
| 5. | ASSESSME | NT OF SAFETY | 76 |
| | 5.1 | Safety Plan | 76 |
| | 5.1.1<br>Emtansine | Risks Associated with Trastuzumab 76 | |
| | 5.1.1.1 | Cardiotoxicity | 77 |
| | 5.1.1.2 | Hematologic Toxicity (Thrombocytopenia) | 77 |
| | 5.1.1.3 | Hepatotoxicity | 77 |
| | 5.1.1.4 | Pulmonary Toxicity | 78 |
| | 5.1.1.5 | Infusion-related Reactions/Hypersensitivity | 78 |
| | 5.1.1.6 | Neurotoxicity | 79 |
| | 5.1.1.7 | Extravasation | 79 |
| | 5.1.1.8 | Trastuzumab Emtansine Dose Modification | 79 |
| | 5.1.2 | Risks Associated with Capecitabine | 79 |
| | 5.1.3<br>Emtansine | Risks Associated with Trastuzumab and Capecitabine Combination | 81 |
| | 5.1.4 | Definition of Dose-limiting Toxicity | 81 |
| | | nsine—F. Hoffmann-La Roche Ltd<br>/ersion 4, 23 Mar 2016 | 5 |

| 5.1.5 | Management of Specific Adverse Events | 82 |
|---|---|---|
| 5.1.5.1 | Trastuzumab Emtansine Dose Modification | 82 |
| | .5.1.1 Trastuzumab Emtansine Dose | 0.4 |
| | dification for Thrombocytopenia | 84 |
| | .5.1.2 Trastuzumab Emtansine Dose dification for Hepatotoxicity | 85 |
| | 5.1.2.1 Concurrent elevations of ALT/AST and bilirubin meeting | • |
| | / laboratory criteria | |
| 5.1.: | 5.1.2.3 Transaminase elevations or bilirubin elevation requiring do | |
| • | stment 85<br>.5.1.3 Trastuzumab Emtansine Dose | |
| | dification for Neurotoxicity | 86 |
| | .5.1.4 Trastuzumab Emtansine Dose | 00 |
| | dification for Cardiotoxicity | 86 |
| | .5.1.5 Trastuzumab Emtansine Dose dification/Management for Infusion-related | |
| Rea | actions, Hypersensitivity Reactions | 87 |
| | .5.1.6 Trastuzumab Emtansine Dose dification for Pulmonary Toxicity | 88 |
| | .5.1.7 Trastuzumab Emtansine Dose | |
| | dification for Extravasation | |
| | Capecitabine Dosage Modification | |
| 5.2 | Safety Parameters and Definitions | |
| 5.2.1 | Adverse Events | 89 |
| 5.2.2<br>Reportable | Serious Adverse Events (Immediately e to the Sponsor) | 90 |
| 5.2.3 | | |
| | on-Serious Expedited Adverse Events | |
| 5.2.4 | Pregnancy and Contraception | 91 |
| 5.3 | Methods and Timing for Capturing and Assessing Safety Parameters | 93 |
| 5.3.1 | Adverse Event Reporting Period | 94 |
| 5.3.2 | Eliciting Adverse Event Information | 94 |
| 5.3.3 | Assessment of Severity of Adverse Events | 94 |
| 5.3.4 | Assessment of Causality of Adverse Events | 95 |
| 5.3.5 | Procedures for Recording Adverse Events | 96 |
| 5.3.5.1 | Diagnosis <i>versus</i> Signs and Symptoms | 97 |
| 5.3.5.2<br>Other I | Adverse Events Occurring Secondary to Events | 97 |

**Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 4, 23 Mar 2016

7

| | 5.3.5 | .3 Persistent or Recurrent Adverse Events | 97 |
|---|---|---|---|
| | 5.3.5 | .4 Abnormal Laboratory Values | 98 |
| | 5.3.5 | .5 Abnormal Vital Sign Values | 98 |
| | 5.3.5 | .6 Abnormal Liver Function Tests | 99 |
| | 5.3.5 | .7 Deaths | 99 |
| | 5.3.5 | .8 Pre-Existing Medical Conditions | 100 |
| | 5.3.5 | .9 Lack of Efficacy or Clinical Worsening | 100 |
| | 5.3.5 | .10 Hospitalization or Prolonged Hospitalization | 100 |
| | 5.3.5<br>Over | .11 Adverse Events Associated with an dose or Error in Drug Administration | 100 |
| | 5.4 | Immediate Reporting Requirements from Investigator to the Sponsor | 101 |
| | 5.4.1 | Emergency Medical Contacts | 101 |
| | 5.4.2<br>Events a<br>Interest | Reporting Requirements for Serious Adverse and Non-serious Adverse Events of Special 101 | |
| | 5.4.3 | Reporting Requirements for Pregnancies | 102 |
| | 5.4.3 | .1 Pregnancies in Female Patients | 102 |
| | 5.4.3<br>Patie | .2 Pregnancies in Female Partners of Male ents 102 | |
| | 5.4.3 | .3 Abortions | 103 |
| | 5.4.3 | .4 Congenital Anomalies/Birth Defects | 103 |
| | 5.5 | Follow-up of Patients after Adverse Events | 103 |
| | 5.5.1 | Investigator Follow-up | 103 |
| | 5.5.2 | Sponsor Follow-up | 104 |
| | 5.6 | Post-study Adverse Events | 104 |
| | 5.7 | Expedited Reporting to Health Authorities, Investigators, Institutional Review Boards, and Ethics Committees | 104 |
| 6. | STATISTIC | CAL CONSIDERATIONS AND ANALYSIS PLAN | 105 |
| | 6.1 | Determination of Sample Size | 105 |
| | 6.2 | Summaries of Conduct of Study | |
| | 6.3 | Summaries of Treatment Group Comparability | 107 |
| | 6.4 | Efficacy Analyses | 108 |
| | 6.4.1 | Primary Efficacy Endpoint | |
| | 6.4.2 | Secondary Efficacy Endpoints | 110 |
| | 6.5 | Safety Analyses | 111 |
| Tras | stuzumab Em | tansine—F. Hoffmann-La Roche Ltd | |

Protocol MO28230, Version 4, 23 Mar 2016
| | 6.6 | Pharmacodynamic Analyses | 113 |
|---|---|---|---|
| | 6.7 | Pharmacokinetic Analyses | 113 |
| | 6.8 | Exploratory Analyses | 114 |
| | 6.9 | Interim Analyses | 114 |
| 7. | DATA COLLECTION AND MANAGEMENT | | |
| | 7.1 | Data Quality Assurance | 115 |
| | 7.2 | Electronic Case Report Forms | 115 |
| | 7.3 | Source Data Documentation | 115 |
| | 7.4 | Use of Computerized Systems | 116 |
| | 7.5 | Retention of Records | 116 |
| 8. | ETHICA | AL CONSIDERATIONS | 117 |
| | 8.1 | Compliance with Laws and Regulations | 117 |
| | 8.2 | Informed Consent | 117 |
| | 8.3 | Institutional Review Board or Ethics Committee | 118 |
| | 8.4 | Confidentiality | 118 |
| | 8.5 | Financial Disclosure | 119 |
| 9. | | DOCUMENTATION, MONITORING, AND | 119 |
| | 9.1 | Study Documentation | |
| | 9.2 | Site Inspections | |
| | 9.3 | Administrative Structure | |
| | 9.4 | Publication of Data and Protection of Trade Secrets | |
| | 9.5 | Protocol Amendments | |
| 10. | REFER | ENCES | 121 |
| | | LIST OF TABLES | |
| Tab | ole 1 | Cycle 1 Mean (s.d.) Pharmacokinetic Parameters for Trastuzumab Emtansine Following Trastuzumab Emtansine Administration q3w and qw in Study | 0- |
| Table 2 | | TDM3569g Dose Reduction for Trastuzumab Emtansine (Patients | |
| T-1- | do 2 | | 83 |
| | | Dose Reductions for Trastuzumab Emtansine (Patients with mGC) | 84 |
| | | Emtansine—F. Hoffmann-La Roche Ltd<br>3230, Version 4, 23 Mar 2016 | 8 |

| Table 4 | Trastuzumab Emtansine Dose Modification: Total Serum Bilirubin | |
|---|---|---|
| Table 5 | Trastuzumab Emtansine Dose Modification: Serum ALT or AST | |
| Table 6 | Adverse Event Severity Grading Scale | 95 |
| Table 7 | Guidance for Causal Attribution of Adverse | |
| | Event/Serious Adverse Event | 96 |
| | LIST OF FIGURES | |
| Figure 1 | Molecular Structure of Trastuzumab Emtansine | |
| Figure 2 | MMTV HER2 Fo5 Mammary Tumor Transplants | 41 |
| Figure 3 | Anti-tumor Activity of Trastuzumab Emtansine in | |
| | Combination with Capecitabine in NCI-N87 | |
| Figure 4 | Overview of Study Design | 47 |
| Figure 5 | Overview of Phase I Dose Finding Study Design | 48 |
| Figure 6 | Algorithm for Continuation and Discontinuation of | |
| | Trastuzumab Emtansine Based on Left Ventricular Ejection Fraction Assessments in Patients | 07 |
| | LIST OF APPENDICES | |
| Appendix 1 | Schedule of Assessments | 126 |
| Appendix 2 | Pharmacokinetic Sampling for Phase I, tic Breast and Gastric Cancer Patients | 136 |
| Metasta | tic breast and Gastine Cancer Fatients | 130 |
| Appendix 3 | Response Evaluation Criteria in Solid Tumors | |
| (RECIS | Γ): Modified Excerpt from Original Publication | 138 |
| Appendix 4 | Instructions for Scans in the Event of Isotope | 450 |
| Shortage | e | 150 |
| Appendix 5 | New York Heart Association Classification of | |
| • • | nal Cardiac Capacity | 15 |
| Appendix 6 | ECOG Performance Status | 152 |

# PROTOCOL ACCEPTANCE FORM

TITLE: PHASE I STUDY OF THE COMBINATION OF TRASTUZUMAB **EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE** METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED OR METASTATIC GASTRIC CANCER PATIENTS, FOLLOWED BY A RANDOMIZED, OPEN-LABEL PHASE II STUDY OF TRASTUZUMAB EMTANSINE AND CAPECITABINE VERSUS TRASTUZUMAB EMTANSINE ALONE IN HER2-POSITIVE METASTATIC BREAST CANCER

PROTOCOL NUMBER: MO28230 **VERSION NUMBER: 4 EUDRACT NUMBER:** 2012-001547-46 **TEST PRODUCT:** Trastuzumab emtansine (RO5304020) Capecitabine (RO091978) **MEDICAL MONITOR:** SPONSOR: F. Hoffmann-La Roche Ltd I agree to conduct the study in accordance with the current protocol. Principal Investigator's Name (print)

Please return the signed original of this form {as instructed by XX [e.g., your *local study monitor, the CRO]* [or] {to the contact provided below}. Please retain a copy for your study files.

{Name} {Address}

Principal Investigator's Signature

Date

#### **PROTOCOL SYNOPSIS**

TITLE: PHASE I STUDY OF THE COMBINATION OF TRASTUZUMAB EMTANSINE

(T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST
CANCER AND HER2-POSITIVE LOCALLY ADVANCED/METASTATIC GASTRIC
CANCER PATIENTS, FOLLOWED BY A RANDOMIZED, OPEN-LABEL PHASE II
STUDY OF TRASTUZUMAB EMTANSINE AND CAPECITABINE VERSUS

STUDY OF TRASTUZUMAB EMTANSINE AND CAPECITABINE VERSUS TRASTUZUMAB EMTANSINE ALONE IN HER2-POSITIVE METASTATIC

**BREAST CANCER** 


**EUDRACT NUMBER:** 2012-001547-46


Capecitabine (RO091978)

PHASE: I/II

**INDICATION:** HER2-positive metastatic breast cancer or HER2-positive locally

advanced/metastatic gastric cancer

**SPONSOR:** F. Hoffmann-La Roche Ltd

## **Objectives**

Phase I: Maximum Tolerated Dose (MTD) Finding of Trastuzumab Emtansine (T-DM1) and Capecitabine in Metastatic Breast Cancer (mBC)

## Primary Objective

• To determine the MTD of the combination of trastuzumab emtansine and capecitabine in patients with human epidermal growth factor receptor 2 (HER2)-positive mBC

# **Secondary Objectives**

To assess the:

- Pharmacokinetics (PK) of trastuzumab emtansine, capecitabine, and their metabolites
- Safety of the combination of trastuzumab emtansine and capecitabine
- Overall response rate (ORR)

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

**Primary Objective** 

 To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone in patients with HER2-positive mBC, as measured by ORR by Response Evaluation Criteria for Solid Tumors (RECIST) v.1.1 per investigator local assessment

## Secondary Objectives

- To assess the safety profile of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone
- To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone in mBC patients, as measured by:
  - Time to response (TTR)

# Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

- Duration of response (DoR)
- Time to progression (TTP)
- Time to treatment failure (TTF)
- Progression-free survival (PFS)
- Clinical benefit rate (CBR)
- Overall survival (OS)

# Phase I: MTD Finding of Trastuzumab Emtansine and Capecitabine in Locally Advanced/Metastatic Gastric Cancer (LA/mGC)

#### Primary Objective

 To determine the MTD of the combination of trastuzumab emtansine and capecitabine in patients with LA/mGC

#### Secondary Objectives

To assess the:

- PK of trastuzumab emtansine, capecitabine, and their metabolites
- Safety of the combination of trastuzumab emtansine and capecitabine
- ORR

# Study Design

#### **Description of Study**

This is an international, multicenter study.

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with HER2-positive mBC or LA/mGC using a Phase I design, followed by a randomized, open-label Phase II study to explore the efficacy and safety of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone in HER2-positive mBC. Results from the Phase I study in LA/mGC will be used as supporting information for future studies in the indication (see Figure 4 in the protocol).

#### Phase I: MTD Finding, Cohort 1: mBC

Cohort 1 used a 3 plus 3 classical design to determine the MTD of capecitabine in combination with trastuzumab emtansine. Initially the study had a dose escalation design, but following the occurrence of two DLTs at Dose Level 1 (750 mg/m² capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine), the study design was adapted and the dose de-escalated to 700 mg/m² capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine. At this Dose Level there were no DLTs and following review of the safety data, the Independent Data Monitoring Committee (IDMC) recommended that the study should proceed to explore this Dose Level further in the Randomized Phase II part of the study.

## Randomized Phase II: Exploration of Efficacy and Safety in mBC

Phase II will be conducted in mBC patients only. This part of the study will explore the efficacy and safety of the combination treatment of trastuzumab emtansine (T-DM1) and capecitabine, at 700 mg/m² bid (the recommended MTD), compared with trastuzumab emtansine alone in patients with mBC.

Approximately 160 additional patients with HER2-positive mBC will be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to the Phase II part of the study; however, they will be followed up until end of study (EOS).

# Phase I: MTD Finding, Cohort 2: LA/mGC

Cohort 2 will have a 3 plus 3 classical design and enroll patients with HER2-positive LA/mGC. Trastuzumab emtansine will be administered weekly at a dose of 2.4 mg/kg and capecitabine will start at dose level -1 (700 mg/m², the MTD defined in Cohort 1), with de-escalation if required as follows:

- If Dose Level -1 is well tolerated (DLT in ≤ 1/6 patients), this dose will be established as the MTD for LA/mGC
- If Dose Level -1 is not tolerated in Cohort 2 (DLT in > 1/6 patients), de-escalation will be to Dose Level -2.

# Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

 If Dose Level -2 is too toxic, the combination of capecitabine with trastuzumab emtansine 2.4 mg/kg every week may be considered unfeasible in LA/mGC, recruitment will be terminated and the LA/mGC part will be closed. However, this will have no impact on continuation of the Randomized Phase II mBC part.

#### **Duration of treatment and follow-up**

All patients will be treated until investigator-assessed disease progression, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor. In case of toxicities requiring the discontinuation of capecitabine, single agent trastuzumab emtansine may be continued. In case of toxicities requiring the discontinuation of trastuzumab emtansine, the patient will be followed up until EOS (treatment with capecitabine alone is not allowed).

All patients will be followed up until withdrawal of consent, death, or for up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first

#### **Number of Patients**

Phase I, Cohort 1: mBC

A minimum of 6 and up to 18 patients will be enrolled.

Randomized Phase II: Exploration of Efficacy and Safety in mBC

Exploration of efficacy and safety in mBC will be based on approximately 160 randomized patients in total.

Phase I, Cohort 2: LA/mGC

A total of 6 to 12 patients will be enrolled.

#### **Target Population**

Phase I, Cohort 1: mBC

Patients with HER2-positive mBC will be enrolled.

The patient's HER2 status will be considered positive if the local institution or reference lab reported immunohistochemistry (IHC) 3+ staining intensity (on a scale of 0 to 3) or *in situ* hybridization (ISH) positive.

The HER2 status will be retrospectively confirmed by IHC and/or ISH in a central laboratory using archival paraffin-embedded tumor tissue. Retrospective central confirmation will not affect the treatment decisions or primary endpoint of Phase I and will be used to validate efficacy analyses in Phase I.

Before entering the study, patients must have received at least one prior treatment regimen for early or metastatic disease, which included a chemotherapy agent and trastuzumab either separately or in combination.

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

Patients with HER2-positive mBC will be randomized to receive either the combination of trastuzumab emtansine with capecitabine or trastuzumab emtansine alone. Retrospective central confirmation will be used to categorize patients for subgroup analyses according to central HER2 testing.

Before entering the study, patients must have received at least one prior treatment regimen for early or metastatic disease, which included a chemotherapy agent and trastuzumab either separately or in combination.

#### Phase I, Cohort 2: LA/mGC

Patients with centrally confirmed HER2-positive LA/mGC will be enrolled.

Patients must not have received prior chemotherapy for advanced/metastatic disease.

## Inclusion Criteria:

#### For mBC Patients:

- 1. Male or female.
- 2. Age ≥ 18 years old.
- 3. Signed informed consent before any study-specific procedure.

# Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

- 4. Able and willing to comply with the protocol.
- 5. Negative serum pregnancy test for women of childbearing potential (including premenopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in the medical history confirming that the patient is not of childbearing potential.
- 6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 7 months after the last dose of study treatment (see Section 5.2.4 in the protocol).
- 7. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
- 8. Blood:
  - a) Platelet count > 100,000 cells/mm<sup>3</sup>
  - b) International normalized ratio (INR) < 1.5
  - c) Absolute neutrophil count (ANC) > 1,500 cells/mm<sup>3</sup>
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 9. Liver function:
  - a) Total bilirubin ≤ 1.5 × upper limit of normal (ULN) or direct bilirubin ≤ 1.5 × ULN in patients with documented Gilbert's syndrome.
  - b) Serum glutamic oxaloacetic transaminase (SGOT)/aspartate transaminase (AST) and serum glutamic pyruvic transaminase (SGPT)/alanine transaminase (ALT) ≤ 2.5 × ULN.
  - c) Alkaline phosphatase  $\leq$  2.5 × ULN. In patients with bone metastases: alkaline phosphatase  $\leq$  5 × ULN.
  - d) Evidence of stable liver function during the month prior to enrollment with liver function test (LFT) fluctuations not exceeding 2.5 × ULN (for AST, ALT) and 1.5 × ULN (for total bilirubin).
- 10. Renal function:
  - a) Serum creatinine of < 177 μmol/L or calculated creatinine clearance (CL)</li>
     > 50 mL/min. If urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate ≤ 1 g of protein/24 hours.
- 11. Cardiac function:
  - a) Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan.
- 12. Life expectancy ≥12 weeks
- 13. Histologically or cytologically confirmed breast cancer.
- 14. HER2-positive disease, defined as IHC 3+ or ISH positive.
- 15. Tumor block or 8 slides available for retrospective central confirmation of HER2-positivity (central confirmation not necessary for enrollment).
- 16. mBC with at least one measurable lesion according to RECIST v.1.1.
- 17. Disease progression on at least one prior regimen containing trastuzumab and chemotherapy either separately or in combination. Patients may be eligible to receive study therapy in the first-line setting if trastuzumab and chemotherapy were given in the [neo]adjuvant setting.
- 18. Patients must have recovered from previous treatments

#### For LA/mGC Patients:

1. Male or female

#### Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

- Age ≥ 18 years old.
- 3. Signed informed consent before any study-specific procedure.
- 4. Able and willing to comply with the protocol.
- 5. Negative serum pregnancy test for women of childbearing potential (including premenopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in the medical history confirming that the patient is not of childbearing potential.
- 6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 7months after the last dose of study treatment (see Section 5.2.4 in the protocol).
- 7. ECOG performance status of 0, 1, or 2.
- 8. Blood:
  - a) Platelet count > 100,000 cells/mm<sup>3</sup>.
  - b) INR < 1.5.
  - c) ANC > 1,500 cells/mm<sup>3</sup>.
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 9. Liver function:
  - a) Total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤ 1.5 × ULN in patients with documented Gilbert's syndrome.
  - b) SGOT/AST and SGPT/ALT ≤ 2.5 × ULN.
  - c) Alkaline phosphatase ≤ 2.5 × ULN. In patients with bone metastases: alkaline phosphatase ≤ 5 × ULN.
  - d) Evidence of stable liver function during the month prior to enrollment with LFT fluctuations not exceeding 2.5 × ULN (for AST, ALT) and 1.5 × ULN (for total bilirubin).
- 10. Renal function:
  - a) Serum creatinine of < 177  $\mu$ mol/L or calculated creatinine CL > 50 mL/min. If urine dipstick for proteinuria is  $\geq$  2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate  $\leq$  1 g of protein/24 hours.
- 11. Cardiac function:
  - a) LVEF ≥ 50% by ECHO or MUGA scan.
- 12. Life expectancy ≥ 2 weeks
- 13. Histologically or cytologically confirmed mGC or locally advanced GC.
- 14. HER2-positive tumor (primary tumor or metastatic lesion), defined as either IHC 3+ or IHC 2+ and ISH+, prospectively confirmed by a Sponsor-designated central laboratory prior to enrollment. ISH positivity is defined as a ratio of ≥ 2.0 for the number of HER2 gene copies to the number of signals for CEP17.
  - a) Archival tumor samples obtained from primary or metastatic sites are acceptable.
  - b) Invasive tumor for central confirmation of HER2 status is required.
  - c) A formalin-fixed paraffin-embedded (FFPE) tissue block with at least 5 mm of invasive tumor for central confirmation is preferred. If FFPE tissue blocks (or partial block) are unavailable due to country or site regulations, a minimum of 8 freshly cut unstained slides MUST be available for central review of HER2 status.
- 15. Inoperable LA/mGC.

## **Exclusion Criteria:**

# For mBC Patients:

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or five half-lives, whichever is longer.
  - b) Hormonal therapy within 14 days.
  - c) Trastuzumab within 21 days.
- 2. Prior treatment with trastuzumab emtansine or prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine.
- 3. Prior treatment with capecitabine.
- History of severe or unexpected reactions to fluoropyrimidine or known hypersensitivity to fluorouracil.
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogs, such as brivudine.
  - b) Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
  - c) Known complete absence of dihydropyrimidine dehydrogenase (DPD) activity.
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product.
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>.
  - b) Epirubicin > 900 mg/m<sup>2</sup>.
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control symptoms within 28 days before first study drug administration.
- 9. Current peripheral neuropathy of Grade ≥ 3 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.4.0.
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above.
- 11. Current unstable ventricular arrhythmia requiring treatment.
- 12. History of symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] Classes II–IV).
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration.
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment.
- 15. Severe dyspnea at rest due to complications of advanced malignancy or currently requiring continuous oxygen therapy.
- 16. Clinically significant malabsorption syndrome or inability to take oral medication.
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease).
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment.
- 19. Current pregnancy or lactation.

#### Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

- 20. Current known active infection with human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C virus (HBV/HCV).
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV deoxyribonucleic acid (DNA) viral load per local guidelines.
- 21. Lapatinib ≤ 14 days before first study drug administration.
- 22. Previous radiotherapy for the treatment of mBC is not allowed if:
  - a) The last fraction of radiotherapy has been administered within 14 days prior to first study drug administration (28 days for patients with radiotherapy to control symptoms of brain metastases, see exclusion criterion 8).
  - b) More than 25% of marrow-bearing bone has been irradiated.
  - c) Any acute toxicity has not resolved to Grade ≤ 1 before first study drug administration.

#### For LA/mGC Patients:

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half-lives, whichever is longer.
  - b) Hormonal therapy within 14 days.
  - c) Trastuzumab within 21 days.
- 2. Prior treatment with trastuzumab emtansine or prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine.
- 3. Prior treatment with capecitabine.
- History of severe or unexpected reactions to fluoropyrimidine or known hypersensitivity to fluorouracil.
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogs, such as brivudine.
  - b) Rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucosegalactose malabsorption.
  - c) Known complete absence of DPD activity.
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product.
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>.
  - b) Epirubicin > 900 mg/m<sup>2</sup>.
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>.
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m² doxorubicin.
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control symptoms within 28 days before first study drug administration.
- 9. Current peripheral neuropathy of Grade ≥ 3 according to NCI CTCAE, v4.0.
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above.
- 11. Current unstable ventricular arrhythmia requiring treatment.
- 12. History of symptomatic CHF (NYHA Classes II-IV).
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration.
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment.

# Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

- 15. Severe dyspnea at rest due to complications of advanced malignancy or currently requiring continuous oxygen therapy.
- 16. Clinically significant malabsorption syndrome or inability to take oral medication.
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation.
- 20. Current known active infection with HIV, HBV, and/or HCV
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Previous chemotherapy for advanced/metastatic disease
  - a) Prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrollment into the study
- 22. Lapatinib ≤ 14 days before first study drug administration

#### Length of Study

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to last 2 years in total (1 year for MTD Finding, 1 year for the Phase II Exploration of Efficacy and Safety in mBC).

# **End of Study**

The study will end after the follow-up period has been completed as defined above. Last patient last visit (LPLV) is defined as the last data collection point, which can be either a clinic visit or a laboratory sample.

In case Dose Level -2 is too toxic in LA/mGC, the LA/mGC cohort may be terminated prematurely. Patients who, at that point, experience response according to RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent or with capecitabine, based on the risk-benefit balance and agreement with the SC.

Randomized Phase II Exploration of Efficacy and Safety in mBC: The primary analysis of best overall response (BOR) rate will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever occurs first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after randomization of the first patient. The EOS analysis (approximately 24 months after the last patient is randomized) will include an updated analysis of BOR, which will be done in a purely exploratory manner.

#### **Efficacy Outcome Measures**

Efficacy will be evaluated according to RECIST v.1.1.

- BOR rate
- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

#### **Safety Outcome Measures**

 DLT assessment/determination of the MTD of capecitabine when combined with trastuzumab emtansine (Phase I only)

#### Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

- Fatal AEs and their causes
- Events to monitor
- Laboratory parameters
- LVEF
- Treatment exposure
- Physical examinations
- ECOG performance status
- Premature withdrawal from study medication and/or study

treatment, and AEs of special interest (AESIs)

## **Pharmacodynamic Outcome Measures**

Hospital visit parameters.

#### **Pharmacokinetic Outcome Measures**

PK will be evaluated during Phase I for trastuzumab emtansine, capecitabine, and their metabolites (see Appendix 1, Schedule of Assessment in the protocol). In addition, PK samples may be taken *ad hoc*, in case of SAEs or unexpected toxicities, which may be suggestive of a potential drug-drug interaction.

### **Investigational Medicinal Products**

#### For mBC Patients:

Trastuzumab emtansine will be administered q3w at a dose of 3.6 mg/kg intravenous (IV).

The total trastuzumab emtansine dose will be calculated based on the patient's weight on Day of each cycle (or up to 3 days before) with no upper limit.

<u>Capecitabine</u> will be administered orally bid for 14 days followed by a 7-day rest period at the Dose Levels described in the 'Trial Design' section.

Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Rounding of the capecitabine dose, based on 150 mg and 500 mg tablet strength, will be allowed to the nearest target dose based on the patient's body surface area (BSA).

#### For LA/mGC Patients:

<u>Trastuzumab emtansine</u> will be administered on Day 1 of each 1-week cycle at a dose of 2.4 mg/kg IV.

The total trastuzumab emtansine dose will be calculated based on the patient's weight on Day of each cycle (or up to 3 days before) with no upper limit.

<u>Capecitabine</u> will be administered orally bid for 14 days followed by a 7-day rest period at the Dose Levels -1 to -2 described in the 'Trial Design' section.

Capecitabine tablets should be swallowed with water within 30 minutes after a meal.

## **Non-Investigational Medicinal Products**

Not applicable.

#### **Statistical Methods**

The study will include 2 phases and 2 cohorts:

- Phase I, Cohort 1: mBC MTD-Finding Cohort
- Randomized Phase II: Exploration of Efficacy and Safety in mBC
- Phase I, Cohort 2: LA/mGC MTD-Finding Cohort

Corresponding analyses as described in the protocol will be performed when all data from both study phases are collected and cleaned.

Randomized Phase II: The primary analysis of BOR will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever occurs first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after

# Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

randomization of the first patient. The EOS analysis (approximately 24 months after the last patient is randomized) will include an updated analysis of BOR, which will be done in a purely exploratory manner.

#### Analysis of primary and secondary endpoints:

#### **Analysis Populations:**

#### Phase I, Cohort 1: MTD-Finding: mBC Patients

The main analysis population for DLT assessment is the DLT-evaluable population, which is defined as all enrolled and treated patients who have not experienced any major protocol violations (including violations of the inclusion and exclusion criteria) and have completed Cycle 1

The safety population (SP) will include all patients who received at least one dose of study medication (trastuzumab emtansine and/or capecitabine) during Phase I.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

The main analysis population for the efficacy analysis will be the intent-to-treat (ITT) population, which will include all patients randomized in the Phase II part of the study. The per-protocol (PP) population will include all ITT patients who have at least one post-baseline tumor assessment during the Phase II part of the study and no major protocol violations, which will be defined in the statistical analysis plan (SAP).

The SP will include all patients who received at least one dose of study medication during the Randomized Phase II part of the study.

#### Phase I, Cohort 2: MTD-Finding, LA/mGC Patients

The main analysis population for DLT assessment is the DLT-evaluable population, which is defined as all enrolled and treated patients who have not experienced any major protocol violation (including violation of the inclusion and exclusion criteria) and have completed Cycle 1.

The SP will include all patients who received at least one dose of study medication during Phase I.

# **Efficacy Endpoints:**

# Phase I, Cohort 1: MTD-Finding, mBC

The primary objectives are defining the MTD and establishing the safety profile of the combination regimen.

ORR, as a main efficacy endpoint, will be assessed via BOR rate. The BOR is defined as the best response recorded from the date of enrollment until disease progression, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

# Randomized Phase II: Exploration of Efficacy in mBC

The primary efficacy endpoint for the Phase II part of the study is the ORR, assessed via the BOR rate. BOR is defined as the best response recorded between randomization into the Phase II part of the study and disease progression, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. To be assigned a status of partial response (PR) or complete response (CR), i.e., to be a responder, changes in tumor measurements must be confirmed by repeated assessments performed no less than 28 days after the response criteria are first met, i.e., patients need to have two consecutive assessments of PR or CR.

The primary hypothesis of interest when comparing ORR – as assessed via BOR - between the two treatment groups, combination of trastuzumab emtansine and capecitabine *versus* trastuzumab emtansine alone is:

#### Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

- H0: π trastuzumab emtansine = π trastuzumab emtansine + capecitabine where π trastuzumab emtansine is BOR in trastuzumab emtansine alone and trastuzumab emtansine + capecitabine is BOR in trastuzumab emtansine + capecitabine
- H: trastuzumab emtansine trastuzumab emtansine + capecitabine

The number and proportions of responders and non-responders (based on BOR) together with the two-sided 90% Clopper-Pearson confidence intervals (CIs) will be presented for each treatment group. The difference in BOR between treatment groups will be displayed with associated 90% CIs using the Hauck-Anderson approach and p-value for the Fisher's exact test.

The secondary endpoints for the Phase II part of the study will be:

- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

Estimates for the survivor function of both treatment groups for TTR, DoR, TTP, TTF, PFS and OS will be obtained by using the Kaplan-Meier method. Hazard ratios and associated 90% CIs will be estimated from non-stratified and stratified (based on the stratification factor) Cox regression models.

CBR will include patients whose best (confirmed) response was PR or CR, or stable disease (SD) that lasted at least 6 months. CBR will be summarized in a similar way to the primary efficacy endpoint, ORR, as assessed by BOR.

## Phase I, Cohort 2: MTD-Finding: LA/mGC

The primary objectives are defining the MTD and establishing the safety profile of the combination regimen.

Efficacy endpoints will be analyzed in a similar way to that described for Phase I, Cohort 1 in mBC.

#### Safety Endpoints:

## Phase I, Cohort 1: MTD-Finding: mBC

The number and proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

Safety parameters for this study part will also be summarized by treatment dose. The summaries of AEs, SAEs, AEs that cause discontinuation from the study treatment, AESIs (as described in Section 5), and events to monitor will be analyzed in a similar way to AEs in Phase II. The summaries will include all patients who received at least one dose of study medication.

The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry will be presented in shift tables of NCI CTCAE grade at baseline *versus* worst grade during treatment for Phase I, Cohort 1.

LVEF over time will be summarized as mean, median and range (minimum and maximum) and will be presented graphically.

Other safety variables, such as exposure to study medication, concomitant medications, and physical examinations, will be analyzed in a similar way. Exposure to study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in each category will be presented by bar charts at different time points.

# Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

## Randomized Phase II: Exploration of Safety in mBC

Safety endpoints will be summarized by treatment group.

Safety endpoints during the Randomized Phase II part of the study will be assessed via: total AEs, Grade ≥ 3 AEs, SAEs, premature withdrawal from study medication, AESIs, events to monitor, laboratory parameters, LVEF, exposure to study medication, concomitant medications, ECOG performance status, and physical examination.

The incidence of AEs and SAEs will be summarized according to the primary SOC and within each SOC, by MedDRA preferred term. Time to onset of the first episode of AESI will also be summarized via Kaplan-Meier method. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology, and biochemistry will be presented in shift tables of NCI CTCAE grade at baseline *versus* worst grade during treatment in the Randomized Phase II part of the study.

LVEF over time will be summarized as mean, median and range (minimum and maximum) and will be presented graphically.

Other safety variables, such as exposure to study medication, concomitant medications, and physical examinations, will be analyzed in a similar way. Exposure to study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in each category will be presented by bar charts at different time points.

#### Phase I, Cohort 2: MTD-Finding: mGC

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

Safety parameters will be summarized in a similar way to that described for Phase I, Cohort 1 in mBC.

#### Pharmacokinetic Analysis

The following PK parameters of trastuzumab emtansine and capecitabine (not limited to these listed) will be determined only in the Phase I part of the study in all patients who receive study treatment using either non-compartmental and/or population methods, if data allow:

- Serum concentrations of trastuzumab emtansine (conjugate) and total trastuzumab
- Plasma concentrations of DM1, capecitabine, and its active metabolite 5-fluorouracil (5-FU)
- Total exposure (area under the serum concentration-time curve [AUC])
- Maximum concentration (C<sub>max</sub>)
- CL
- Volume of distribution (V<sub>d</sub>)
- Terminal half-life (T<sub>1/2</sub>)

All PK parameters will be listed and tabulated by treatment dose and by Cohort. Descriptive summary statistics including arithmetic mean, geometric mean (e.g., AUC and  $C_{max}$ ), median, range, standard deviation (s.d.), and coefficient of variation will be presented for each Cohort. Nonlinear mixed effects modeling will also be used; details will be presented in the SAP.

## **Exploratory Analyses**

For all patients with mBC (Phase I, cohort 1; Phase II Exploration of Efficacy and Safety in mBC), a retrospective central confirmation of the HER2 status will be done. Further exploratory analyses will be done according to centrally confirmed HER2 status for selected endpoints, e.g. BOR and safety (AEs, SAEs, Grade ≥ 3 AEs, and AESIs).

Subgroup analysis for BOR, safety (AEs, SAEs, AEs with Grade ≥ 3, and AESIs) in the Randomized Phase II part of the study will be presented for both treatment groups with respect to: elderly *versus* younger patients; patients with ECOG 0–1 *versus* ECOG 2; and patients with

# Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

≤1 *versus* >1 prior treatment line for metastatic disease. More details will be presented in the SAP.

#### **Pharmacoeconomic Endpoint**

The number of hospital visits, number of days admitted, and type of visits (emergency department *versus* inpatient care) will be collected and compared. The reason for admission (disease progression *versus* AE) will also be assessed.

#### **Determination of Sample Size**

#### Sample Size for Phase I: MTD-Finding: mBC

This part will be based on a classical 3 plus 3 Phase I design. A minimum of 6 and up to 18 patients will be enrolled in Cohort 1. There is no formal sample size estimation for this part.

#### Sample Size for Randomized Phase II: Exploration of Efficacy and Safety in mBC

The sample size for the primary endpoint BOR is based on a Fisher's exact test with an alpha level of 5% (one-sided), power of 70% and the clinical assumption of a BOR rate of 43% with trastuzumab emtansine alone and 62.5% with the combination of trastuzumab emtansine and capecitabine. Approximately 160 patients (approximately 80 patients in each treatment group), including a 15% withdrawal rate, will be randomized with a 1:1 ratio to either trastuzumab emtansine alone or the combination of trastuzumab emtansine and capecitabine.

#### Stratification Factors

The following stratification factor will be implemented in the Randomized Phase II part of the study:

 Number of prior lines of treatment for metastatic disease (≤1 or >1; excluding single-agent hormones).

A treatment line is defined as any treatment regimen given to a patient from treatment initiation until confirmed disease progression.

# Sample Size for Phase I, Cohort 2: MTD-Finding: LA/mGC

This part will be based on a classical 3 plus 3 Phase I design. Between 3 and 12 patients might be enrolled in Cohort 2. There is no formal sample size estimation for this part.

#### Interim analysis

There is no formal interim analysis of efficacy.

An independent data monitoring committee (IDMC) will recommend whether the Randomized Phase II part of the study can commence.

The IDMC will also monitor safety outcomes after 25, 75, and 150 patients have received at least 3 cycles of treatment (Cycle 3 Day 21) in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II part of the study or as requested.

Efficacy data will be provided only if required by the IDMC to estimate the risk-benefit balance for the patients. Further details on the function and logistics of the IDMC will be provided in the IDMC Charter.

# **LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS**

| Abbreviation | Definition |
|---|---|
| ADL | activities of daily living |
| ADC | antibody-drug conjugate |
| AE | adverse event |
| AESI | adverse event of special interest |
| ALT | alanine transaminase |
| ANC | absolute neutrophil count |
| aPTT | activated partial thromboplastin time |
| ARDS | acute respiratory distress syndrome |
| AST | aspartate transaminase |
| AUC | area under the serum concentration-time curve |
| BC | breast cancer |
| bid | twice daily |
| BML | below measurable limit |
| BOR | best overall response |
| BSA | body surface area |
| BUN | blood urea nitrogen |
| CBR | clinical benefit rate |
| CHF | congestive heart failure |
| CI | confidence interval |
| CL | clearance |
| C <sub>max</sub> | maximum concentration |
| CR | complete response |
| CRO | contract research organization |
| CSR | clinical study report |
| CT | computed tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DLT | dose-limiting toxicity |
| DM1 | derivative of maytansine |
| DoR | duration of response |
| DPD | dihydropyrimidine dehydrogenase |
| DPYD | dihydropyrimidine dehydrogenase gene |
| 5-DFUR | 5'-deoxy-5-fluorouridine |
| 5-FU | 5-fluorouracil |
| EC | Ethics Committee |
| ECG | electrocardiogram |
| ECHO | echocardiogram |

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

| ECOG | Eastern Cooperative Oncology Group |
|----------|-------------------------------------------------------------|
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| EEA | European economic area |
| EOS | end of study |
| EU | European Union |
| FDA | Food and Drug Administration |
| FFPE | formalin-fixed paraffin-embedded |
| FISH | fluorescence in situ hybridization |
| GC | gastric cancer |
| GCP | Good Clinical Practice |
| GEJ | gastroesophageal junction |
| HBV | hepatitis B virus |
| HCV | hepatitis C virus |
| HER | human epidermal growth factor receptor |
| HER2 | human epidermal growth factor receptor 2 |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | human immunodeficiency virus |
| HR | hazard ratio |
| ICH | International Conference on Harmonisation |
| IDMC | independent data monitoring committee |
| IgG | immunoglobulin |
| IHC | immunohistochemistry |
| ILD | interstitial lung disease |
| IMP | investigational medicinal product |
| IND | Investigational New Drug (application) |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| ISH | in situ hybridization |
| ITT | intent-to-treat |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| IxRS | interactive voice/web recognition system |
| LA/mGC | locally advanced/metastatic gastric cancer |
| LC-MS/MS | liquid chromatography electrospray tandem mass spectrometry |
| LFT | liver function test |
| LPLV | last patient last visit |

**LVEF** 

SAE

SAP

SC

s.d.

SD

SDV

**SGPT** 

**SmPC** 

SOC

**SWFI** 

T<sub>1/2</sub>

SP

**SGOT** 

| | • |
|--------|---------------------------------------------------------------|
| mBC | metastatic breast cancer |
| mGC | metastatic gastric cancer |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | magnetic resonance imaging |
| MTD | maximum tolerated dose |
| MUGA | multiple-gated acquisition |
| N | number of patients |
| NCI | National Cancer Institute |
| NE | not evaluable |
| NRH | nodular regenerative hyperplasia |
| NYHA | New York Heart Association |
| ORR | overall response rate |
| OS | overall survival |
| PD | progressive disease |
| PET | positron emission tomography |
| PFS | progression-free survival |
| PK | pharmacokinetic |
| PP | per-protocol |
| PR | partial response |
| PVC | polyvinyl chloride |
| QTcF | heart rate-corrected QT interval using the Fridericia formula |
| q3w | every 3 weeks |
| qw | weekly |
| RECIST | Response Evaluation Criteria for Solid Tumors |

serious adverse event

statistical analysis plan

source data verification

system-organ class

sterile water for injection

safety population

terminal half-life

Steering Committee

standard deviation

stable disease

serum glutamic oxaloacetic transaminase

serum glutamic pyruvic transaminase

**Summary of Product Characteristics** 

left ventricular ejection fraction

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

| TTF time to treatment failure | |
|-------------------------------|----------------------------------------|
| TTP | time to progression |
| TTR | time to response |
| ULN | upper limit of normal |
| V <sub>d</sub> | volume of distribution |
| V <sub>ss</sub> | volume of distribution at steady state |
| WBC | white blood cells |
| WHO | World Health Organization |

# 1. <u>BACKGROUND</u>

# 1.1 BACKGROUND ON DISEASE

# 1.1.1 HER2-Positive Breast Cancer

Breast cancer (BC) is the most common cancer in women worldwide, both in the developed and the developing world<sup>1</sup>, with an estimated 1.67 million new cases diagnosed in 2012. It is also the leading cause of cancer death in females in less developed regions, accounting for 324,000 deaths (14.3% of all cancer deaths) in 2012, and the second most common cause of cancer death in women in more developed regions (198,000 deaths, 15.4%) after lung cancer.<sup>1</sup> Metastatic breast cancer (mBC) is incurable, with the primary goal of treatment to extend life and palliate symptoms while preserving quality of life.

Human epidermal growth factor receptor 2 (HER2) is an important prognostic factor in BC and is a key factor influence treatment strategies. The human epidermal growth factor receptor (HER) tyrosine kinase receptor family comprises four receptors: HER1, HER2, HER3, and HER4. These receptors are important mediators of cell growth, survival, and differentiation.<sup>2</sup> Activation of HER receptors leads to receptor dimerization and cell signaling through the PI3-kinase/AKT pathway for promotion of tumor cell survival and through the mitogen-activated protein kinase pathway for cellular proliferation.

Overexpression of HER2 is observed in approximately 15–20% of human BCs. Several lines of scientific and clinical evidence support a direct role for HER2 overexpression in the aggressive growth and poor clinical outcomes associated with these tumors.<sup>3</sup> The development of trastuzumab in the 1990s provided women with HER2-overexpressing tumors with a markedly better outcome than was possible with chemotherapy alone. Increases in overall response rate (ORR), response duration, and progression-free survival (PFS) were associated with a 5-month overall survival (OS) advantage when trastuzumab was given in the first-line metastatic setting, as demonstrated in the initial Phase III trial.<sup>4</sup>

For patients with HER2-positive mBC, the combination of anti-HER2 therapy and a taxane is a globally accepted first-line treatment, based on the OS advantage demonstrated in three large pivotal trials.<sup>4–6</sup>

However, disease progresses in almost all patients with HER2-positive mBC and these patients require additional therapies. Importantly, such tumors continue to express high levels of HER2,<sup>7</sup> and neither the process of internalization nor the level of surface expression is altered when HER2 is bound by trastuzumab.<sup>8</sup>

After progression, the standard strategy is further HER2-directed therapy, either continuing trastuzumab with a different chemotherapy agent (eg trastuzumab plus capecitabine), or changing to a different HER2-directed regimen (eg lapatinib plus capecitabine). In a randomized Phase III trial, GBG26, in patients

whose disease had progressed on previous trastuzumab-containing therapy, the combination of trastuzumab and capecitabine was associated with significantly improved time to progression (TTP) (hazard ratio [HR] 0.69, median 8.2 *versus* 5.6 months, respectively) and ORR (48% *versus* 27%) compared with capecitabine alone. In another Phase III trial involving patients with advanced HER2-positive BC previously treated with an anthracycline, a taxane, and trastuzumab, the addition of lapatinib to capecitabine resulted in an increased ORR (24% *versus* 14%) and TTP (median 6.2 months *versus* 4.3 months) compared with capecitabine alone.

# 1.1.2 HER2-Positive Locally Advanced/Metastatic Gastric Cancer

Gastric cancer (GC) remains one of the most common malignancies in the world with an estimated 952,000 new cases in 2012.¹ GC also continues to be a deadly disease; it is the third leading cause of cancer-related death, accounting for 723,000 deaths (8.8% of all cancer deaths) worldwide in 2012. The only potentially curative treatment for GC is complete resection of localized disease. The overall 5-year survival for all cases, regardless of initial stage at diagnosis, is less than 25%.¹¹¹-¹⁴ Among patients with localized disease who undergo curative surgery, approximately 40–60% will have disease recurrence. Patients with unresectable disease due to locally advanced growth or metastatic spread have the poorest prognosis, with an overall 5-year survival rate in the range of 3% to 15%.¹¹¹,¹³,¹⁴

Whereas HER2 overexpression is associated with a poor prognosis in BC, the prognostic significance of HER2 overexpression in GC is not fully defined. Studies of HER2 positivity rates in GC have shown a broad variation of HER2 positivity ranging from 6.8% to 34.0% for immunohistochemistry (IHC) and 7.1% to 42.6% for fluorescence *in situ* hybridization (FISH) techniques. <sup>15,16</sup> In a recent study, HER2 positivity was shown in 17% of resected esophageal adenocarcinomas and was significantly associated with lower tumor grade, less invasiveness, fewer malignant nodes, and the presence of adjacent Barrett's esophagus. <sup>17</sup>

In the ToGA trial (study BO18255), a global, Phase III study of trastuzumab plus chemotherapy as first-line treatment for advanced HER2-positive GC, <sup>18</sup> an overall HER2-positivity rate of 22.1% was observed (810/3667 evaluable samples), which is similar to BC. A higher HER2 positivity rate was seen in adenocarcinoma of the gastroesophageal junction (GEJ) than in the stomach (33.2% *versus* 20.9%), and intestinal type GCs showed a significantly higher HER2 positivity rate than diffuse or mixed-type tumors (intestinal: 32.2%, diffuse: 6.1%, mixed: 20.4%). <sup>19</sup>

In the ToGA trial, the addition of trastuzumab to chemotherapy (capecitabine or fluorouracil combined with cisplatin) for the treatment of patients with HER2-positive (defined as IHC 3+ or FISH positive), inoperable, locally advanced or recurrent and/or metastatic adenocarcinoma of the stomach or GEJ resulted in

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd Protocol MO28230, Version 4, 23 Mar 2016 an increase in OS (median 13.8 months *versus* 11.1 months, HR 0.74, p = 0.0046), ORR (47% *versus* 35%), PFS (median 6.7 *versus* 5.5 months), and TTP (median 7.1 *versus* 5.6 months) compared with chemotherapy alone.<sup>18</sup>

# 1.2 BACKGROUND ON STUDY DRUGS

# 1.2.1 TRASTUZUMAB EMTANSINE

Trastuzumab emtansine (Figure 1) is a novel antibody-drug conjugate (ADC) that is specifically designed for the treatment of HER2-positive malignancies. Trastuzumab emtansine is composed of: trastuzumab, a humanized monoclonal antibody directed against the extracellular region of HER2; an average of 3.5 molecules of derivative of maytansine (DM1; maytansinoid), an anti-microtubule agent; and the thioether linker maleimidylmethyl cylcohexane-1-carboxylate, which is used to conjugate each molecule of DM1 to trastuzumab. DM1 is a highly potent drug synthesized from maytansinol that binds  $\beta$  tubulin to inhibit tubulin polymerization. It binds to tubulin competitively with vinca alkaloids, but is 20–100 times more potent than vincristine in its cytotoxic effect against tumor cell lines. Its parent molecule, maytansine, was studied in approximately 800 cancer patients in the 1970s and 1980s, with responses seen in patients with breast and lung cancers.  $^{20,21}$  However, because of its narrow therapeutic index and the observed gastrointestinal toxicity of the free drug, it was not developed further as a therapeutic option.  $^{22,23}$ 

Figure 1 Molecular Structure of Trastuzumab Emtansine



DM1 = Derivative of maytansine, a microtubule destabilizing agent MW = Molecular weight

Similar to trastuzumab, trastuzumab emtansine recognizes an epitope in the extracellular domain of HER2 and binds to HER2 with a similar affinity. Following antigen-specific binding of trastuzumab emtansine to HER2, the complex of receptor and ADC is internalized, whereupon DM1-containing catabolites are released into the cytosol following proteolytic cleavage of the antibody in lysosomes.  $^{24}$  Binding of these DM1-containing species to  $\beta$ -tubulin inhibits tubulin polymerization, resulting in cell death.  $^{22}$ 

In addition to targeting delivery of DM1 to HER2-overexpressing tumor cells, trastuzumab emtansine retains the anti-tumor activities of trastuzumab, including suppression of HER2 signaling pathways that confer a proliferative and survival advantage to cells, and the flagging of cells for destruction through antibody-dependent cell cytotoxicity.<sup>20</sup>

Phase I single-arm studies were conducted to identify the most appropriate dosing regimen for further clinical development, and assess the safety of trastuzumab emtansine. Low levels of DM1 in systemic circulation supported the stability of the linker. The studies also provided an indication of clinical activity and led to randomized evaluation of single-agent trastuzumab emtansine versus other HER2-directed therapy in combination with chemotherapy. These trials demonstrated significantly superior PFS and OS with trastuzumab emtansine. English emansion of the safety of trastuzumab emtansine and the safety of trastuzumab emtansine versus other HER2-directed therapy in combination with chemotherapy. These trials demonstrated significantly superior PFS and OS with trastuzumab emtansine.

Data from clinical trials of trastuzumab emtansine that are relevant to the design of the current trial are summarized below. Please refer to the trastuzumab emtansine Investigator's Brochure for further information on all of the completed and ongoing trastuzumab emtansine studies.

# 1.2.1.1 Study TDM3569g

Study TDM3569g was a Phase I, dose-escalation study that evaluated the safety and efficacy of trastuzumab emtansine as a single agent in 52 patients with HER2-positive mBC, whose disease progressed on a trastuzumab-containing chemotherapy regimen.<sup>29,30</sup> The study was completed on 11 June 2009, with a total of 52 patients treated; 24 patients received trastuzumab emtansine every 3 weeks (q3w); 28 patients received trastuzumab emtansine on a weekly (qw) schedule.

On the q3w dosing schedule, dose-limiting toxicities (DLTs) of Grade 4 thrombocytopenia were seen in 2 of 3 patients treated at 4.8 mg/kg. Therefore, 3.6 mg/kg was determined to be the maximum tolerated dose (MTD) of trastuzumab emtansine given q3w, and the cohort was expanded to 15 patients. On the basis of these data, the recommended dose schedule for the Phase II studies was 3.6 mg/kg q3w. On the qw schedule, 2.4 mg/kg was identified as the MTD.

Treatment with trastuzumab emtansine was well tolerated, and toxicity was generally mild, reversible, and non-cumulative. No drug-related cardiac toxicity was noted.

Trastuzumab emtansine administration demonstrated considerable activity in this Phase I study. The confirmed ORR in patients with measurable disease at the 3.6 mg/kg q3w schedule was 44% (4 of 9 patients), as assessed by investigators. The median PFS among the 15 patients receiving 3.6 mg/kg q3w was 10.4 months.

# 1.2.1.2 Study TDM4258g

Study TDM4258g was a Phase II study that evaluated the safety and efficacy of trastuzumab emtansine administered at a dose of 3.6 mg/kg (intravenous; IV) q3w in patients with HER2-positive mBC whose disease had progressed on previous HER2-directed therapy and conventional chemotherapy.<sup>31</sup>

The primary objectives for this study were: 1) to assess the ORR (by independent radiologic review) associated with trastuzumab emtansine 3.6 mg/kg IV q3w; and 2) to characterize the safety and tolerability of trastuzumab emtansine at this dose.

The study was activated on 20 July 2007, and enrollment was completed (n = 112) on 31 July 2008. The final analysis of ORR was performed with a data cut-off date of 25 June 2009, 11 months after the last patient was enrolled. The reported ORR in all patients was 37.5% (95% confidence interval [CI]: 28.6%—

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd Protocol MO28230, Version 4, 23 Mar 2016 46.6%) by investigator assessment and 25.9% (95% CI: 18.4%–34.4%) by independent review. The clinical benefit rate (CBR; defined as complete response [CR], partial response [PR], or stable disease [SD] for >6 months) was 46.3% by investigator assessment and 39.3% by independent review. The median PFS was 4.6 months as assessed by both the investigators and independent review. In the subset of patients whose archival primary tumors were retrospectively confirmed to be HER2-positive (74 of 95 patients with submitted tumor samples), the ORR was 33.8% by independent review and 47.3% based on investigator assessment.

The most common adverse events (AEs) (occurring in  $\geq$  20% of patients) were fatigue (65.2%), nausea (50.9%), headache (40.2%), epistaxis (35.7%), pyrexia (34.8%), constipation (30.4%), cough (27.7%), hypokalemia (26.8%), diarrhea (25.9%), vomiting (24.1%), arthralgia (22.3%), pain in extremity (22.3%), anemia (20.5%), and dyspnea (20.5%). Most of these AEs were Grade 1–2. The three most common Grade 3–4 AEs observed in this trial were hypokalemia (8.9%), thrombocytopenia (8.0%), and fatigue (4.5%). There was one reported Grade 5 event in a patient who died of respiratory failure attributed by the investigator to underlying disease. No Grade  $\geq$  3 left ventricular systolic dysfunction events (symptomatic congestive heart failure [CHF] and/or left ventricular ejection fraction [LVEF] of < 40%) were observed.

# 1.2.1.3 Study TDM4374g

Study TDM4374g was a Phase II, single-arm study of trastuzumab emtansine administered at 3.6 mg/kg by IV infusion q3w to patients with HER2-positive mBC.<sup>32</sup> Patients must have received an anthracycline, trastuzumab, a taxane, lapatinib, and capecitabine given in the neoadjuvant, adjuvant, or metastatic setting or as treatment for locally advanced disease. Patients must have been treated with two HER2-directed therapies in the metastatic or locally advanced setting and have experienced progressive disease (PD) on their most recent treatment.

The primary objectives of this study were: 1) to assess the ORR as determined by an independent review using the modified Response Evaluation Criteria for Solid Tumors (RECIST) v. 1.0; and 2) to characterize the safety and tolerability of this trastuzumab emtansine regimen in the aforementioned patient population. The study was activated on 2 May 2008, and enrollment was complete on 2 April 2009. A total of 110 patients were enrolled and treated in the study.

An efficacy analysis (data cut-off date: 21 June 2010) with a median follow-up of 17.4 months demonstrated an ORR (CR or PR) of 34.5% (95% CI: 26.1%–43.9%; 38 of 110 patients) by independent review and 32.7% (95% CI: 24.1%–42.1%; 36 patients) by investigator assessment. The CBR was 48.2% by independent review and 46.4% by investigator assessment. The median duration of response (DoR) and median PFS by independent review was 7.2 months and 6.9 months, respectively. In the subset of patients whose archival primary tumors were retrospectively confirmed to be HER2-positive (80 of 95 patients with submitted

tumor samples), the ORR was 41.3% by independent review and 40.0% based on investigator assessment.

The most common AEs (occurring in  $\geq$  20% of patients) were fatigue (61.8%), thrombocytopenia (38.2%), nausea (37.3%), increased aspartate transaminase (AST, 26.4%), constipation (23.6%), pyrexia (22.7%), epistaxis (22.7%), headache (21.8%), hypokalemia (20.9%), decreased appetite (20.9%), dry mouth (20.0%), and anemia (20.0%). Most of these AEs were Grade 1–2. Fifty-two patients (47.3%) experienced at least one Grade  $\geq$  3 AE, the most common being thrombocytopenia (9.1%) and fatigue (4.5%). Serious AEs (SAEs) were recorded in 28 patients (25.5%), the most common being cellulitis (3.6%), pyrexia (2.7%), and pneumonia (2.7%). There was one Grade 5 AE (hepatic dysfunction), which was recorded as possibly related to trastuzumab emtansine. The patient had pre-existing non-alcoholic fatty liver disease as well as multiple other comorbidities, including renal insufficiency.

# 1.2.1.4 Study TDM4450g

This was a randomized, multicenter, Phase II study of the efficacy and safety of trastuzumab emtansine *versus* trastuzumab plus docetaxel in patients with metastatic HER2-positive BC who had not received prior chemotherapy for metastatic disease.<sup>26</sup> This study completed enrollment in December 2009 (n = 137). The co-primary objectives were to assess the efficacy of trastuzumab emtansine compared with the combination of trastuzumab and docetaxel, as measured by PFS based on investigator tumor assessments, and to characterize the safety of trastuzumab emtansine compared with the combination of trastuzumab and docetaxel in this population. Secondary endpoints included ORR, OS, and DoR.

The data cut-off date was 15 November 2010. Seventy patients were randomized to the control arm and 67 patients to the trastuzumab emtansine arm. The median duration of follow-up was 13.5 months for the control arm and 13.8 months for the trastuzumab emtansine arm.

As of 15 November 2010, the median PFS was 14.2 months in the trastuzumab emtansine arm versus 9.2 months in the trastuzumab plus docetaxel arm. The HR for PFS was 0.594 (95% CI: 0.364–0.968; p = 0.0353). The ORR in the trastuzumab emtansine arm was 64.2% (95% CI: 51.8%–74.8%) compared with 58.0% (95% CI: 45.5%–69.2%) in the control arm (based on 69 evaluable patients). The CBR was 74.6% (95% CI: 63.2%–84.2%) in the trastuzumab emtansine arm versus 81.2% (95% CI: 70.7%–89.1%) in the trastuzumab plus docetaxel arm (based on 69 evaluable patients). Based on safety data analyzed at the data cut-off date, single-agent trastuzumab emtansine appears to have a favorable overall safety profile compared with trastuzumab and docetaxel as first-line therapy for mBC. The incidence of Grade  $\geq$  3 AEs in the control arm (89.4%; n = 66) was nearly twice that of trastuzumab emtansine (46.4%; n = 69). The rates of SAEs for both arms were similar (control arm 25.8% versus trastuzumab emtansine 18.8%). One patient in the trastuzumab emtansine group died as a

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd Protocol MO28230, Version 4, 23 Mar 2016 result of an AE (sudden death). This patient was randomized to receive trastuzumab plus docetaxel but mistakenly received a single dose of 6 mg/kg trastuzumab emtansine instead of 6 mg/kg trastuzumab. One patient in the trastuzumab plus docetaxel group died due to cardiopulmonary failure. With respect to cardiotoxicity, based on local assessments of LVEF, trastuzumab emtansine was not associated with an increase in cardiotoxicity compared with trastuzumab plus docetaxel.

# 1.2.1.5 Study TDM4688g

The effect of trastuzumab emtansine (3.6 mg/kg q3w) on the QT interval in patients with HER2-positive recurrent locally advanced BC or mBC was evaluated in study TDM4688g. No meaningful effect of trastuzumab emtansine on the corrected QT interval was seen in these patients. At Cycle 1 Day 1, 15 minutes post-infusion, the baseline-adjusted mean heart rate-corrected QT interval using the Fridericia formula (QTcF) increased by 1.2 ms. By 60 minutes post-infusion, the baseline-adjusted mean QTcF interval decreased by 1.0 ms, and by Day 8 of Cycle 1 the baseline-adjusted mean QTcF interval decreased by 4.0 ms. By Cycle 3 Day 1, prior to trastuzumab emtansine infusion, the mean QTcF interval had reverted to baseline. Following the third infusion of trastuzumab emtansine, the baseline-adjusted mean QTcF interval at both the 15-minute and the 60-minute post-infusion time points was increased by 4.7 ms. No patient exhibited a mean change in QTcF interval from baseline exceeding 30 ms at any of the protocol-specified time points.

The relationship between trastuzumab emtansine pharmacokinetic (PK) and electrocardiogram (ECG) data was also assessed. While there appears to be a trend between trastuzumab emtansine drug concentration and its effect on QT interval, at the observed concentration ranges of trastuzumab emtansine, DM1, and total trastuzumab, there is reasonable assurance that the true increase in mean baseline-adjusted average QTcF does not exceed 5 ms. Moreover, because trastuzumab emtansine, total trastuzumab, and DM1 achieve steady state levels by Cycle 3, the likelihood of progressively longer QTcF with repeated trastuzumab emtansine dosing is low.

In this study, the ORR was 25.5% (95% CI: 15.2%–38.5%) as assessed by the investigator; no independent review was performed. The CBR was 39.2% (95% CI: 25.8%–53.1%), and the median PFS was 4.3 months (95% CI: 4.0–6.7).

# 1.2.1.6 Phase III Study TDM4370g

A randomized, open-label Phase III trial (TDM4370g; EMILIA) compared single-agent trastuzumab emtansine *versus* lapatinib and capecitabine in patients with HER2-positive locally advanced unresectable BC or mBC who had received a prior taxane and trastuzumab therapy and had documented PD.<sup>27</sup>

Patients were randomized in a 1:1 ratio to trastuzumab emtansine 3.6 mg/kg IV q3w or the combination of oral capecitabine 1,000 mg/m² twice daily (bid) on

Days 1–14 q3w plus oral lapatinib 1,250 mg/day given as continuous dosing. Treatment was continued until PD (as assessed by the investigator), unmanageable toxicity, or study termination. PFS and OS were co-primary endpoints, with PFS based on modified RECIST<sup>34</sup> and assessed by independent review. Key secondary endpoints were ORR, DoR, and CBR, determined both by the investigator and by independent review.

The study demonstrated statistically significant and clinically meaningful improvements in both PFS and OS for trastuzumab emtansine compared with lapatinib plus capecitabine. Median PFS was 9.6 months in the trastuzumab emtansine arm *versus* 6.4 months in the control arm (HR = 0.65; 95% CI: 0.55–0.77; p < 0.001, log-rank test). Median OS was 30.9 months *versus* 25.1 months, respectively (HR = 0.68; 95% CI: 0.55–0.85; p < 0.001, log-rank test).

This benefit was supported by consistent improvements in all secondary efficacy endpoints, including investigator-assessed PFS, ORR, time to treatment failure (TTF), and the patient-reported outcome of time to symptom progression. The ORR in the trastuzumab emtansine arm was 43.6% (95% CI: 38.6%–48.6%) compared with 30.8% (95% CI: 26.3%–35.7%) in the control arm (based on 786 evaluable patients). Single-agent trastuzumab emtansine appears to have a favorable overall safety profile compared with lapatinib and capecitabine in mBC. The incidence of Grade  $\geq 3$  AEs in the control arm (56.9%; n = 488) was 278; that of trastuzumab emtansine (40.8%; n = 490) was 200. The rates of SAEs for both arms were similar (control arm 18% *versus* trastuzumab emtansine 15.5%).

Based on the results of this phase III trial, both the Food and Drug Administration (FDA) in the US and the European Commission in Europe approved trastuzumab emtansine for the treatment of HER2-positive mBC previously treated with trastuzumab and a taxane.

# 1.2.1.7 Phase III study TDM4997g

A second open-label randomized Phase III trial (TDM4997g; TH3RESA) compared single-agent trastuzumab emtansine *versus* the investigator's choice of therapy in patients with HER2-positive advanced BC who had previously received two or more HER2-directed regimens in the advanced setting, including trastuzumab and lapatinib, and previous taxane therapy in any setting.<sup>28</sup> A total of 602 patients were randomized in a 2:1 ratio (404 to trastuzumab emtansine and 8 to physician's choice).

After median follow-up of approximately 7 months in both arms, 219 patients (54%) in the trastuzumab emtansine group and 2 (65) in the physician's choice group had experienced PFS events. PFS was significantly improved with trastuzumab emtansine compared with physician's choice (HR 0.528, p<0.0001; median PFS 6.2 months with trastuzumab emtansine *versus* 3.3 months in the control arm. The HR for OS at the interim analysis was 0.552 (95% CI 0.369–0.826) but the stopping boundary was not crossed.

Grade ≥3 AEs occurred less frequently with trastuzumab emtansine than with physician's choice (32 of patients vs 43 ). Grade ≥3 neutropenia, diarrhea, and febrile neutropenia were less common with trastuzumab emtansine than physician's choice, whereas grade ≥3 thrombocytopenia (5% vs 2%) was more common with trastuzumab emtansine.

## 1.2.1.8 Pharmacokinetics

The PK of trastuzumab emtansine and its analytes (total trastuzumab and DM1) were characterized in one Phase I study (TDM3569g) and three Phase II studies (TDM4258g, TDM4374g, and TDM4688g).

For study TDM3569g, the final PK parameter estimates based on non-compartmental PK analysis for q3w and qw regimens of trastuzumab emtansine administration are presented in Table 1.

Table 1 Cycle 1 Mean (s.d.) Pharmacokinetic Parameters for Trastuzumab Emtansine Following Trastuzumab Emtansine Administration q3w and qw in Study TDM3569g

| Dose<br>(mg/kg) | No. of<br>Patients | C <sub>max</sub><br>(µg/mL) | AUC <sub>inf</sub><br>(day µg/mL) | T <sub>1/2</sub><br>(day) | $V_d$ (mL/kg) | CL<br>(mL/day/kg) |
|---|---|---|---|---|---|---|
| q3w dosing | | | | | | |
| 0.3 | 3 | 9.6 (1.7) | 14.5 (3.4) | 1.3 (0.2) | 35.7 (7.5) | 21.1 (4.5) |
| 0.6 | 1 | 13.3 | 24.5 | 1.3 | 43.8 | 24.5 |
| 1.2 | 1 | 20.3 | 42.9 | 1.3 | 51.8 | 27.8 |
| 2.4 | 1 | 76.3 | 330.0 | 2.2 | 30.7 | 7.2 |
| 3.6 | 15 | 76.2 (19.1) | 300.3 (65.8) | 3.1 (0.7) | 58.4 (12.4) | 12.7 (3.6) |
| 4.8 | 3 | 130.3 (7.8) | 673.0 (12.2) | 4.1 (0.7) | 41.2 (6.2) | 7.1 (0.1) |
| qw dosing | | | | | | |
| 1.2 | 3 | 29.6 (5.7) | 76.2 (10.4) | 2.3 (0.6) | 47.5 (6.0) | 15.9 (2.4) |
| 1.6 | 3 | 34.3 (4.8) | 130.3 (39.7) | 3.4 (0.8) | 59.8 (16.6) | 13.0 (3.4) |
| 2.0 | 3 | 48.0 (9.6) | 175.0 (41.0) | 3.1 (0.3) | 51.0 (8.1) | 11.8 (2.4) |
| 2.4 | 16 | 54.8 (12.6) | 198.5 (54.5) | 3.3 (1.1) | 55.4 (13.0) | 13.1 (4.1) |
| 2.9 | 3 | 78.1 (33.9) | 212.0 (39.0) | 2.9 (0.5) | 57.7 (2.2) | 14.0 (2.6) |

AUC<sub>inf</sub> = area under the serum concentration-time curve from time 0 extrapolated to infinity;  $C_{max}$  = maximum serum concentration; CL = clearance; s.d. = standard deviation;  $T_{1/2}$  = terminal half-life;  $V_d$  = volume of distribution.

Dose intensity, defined as percentage of the planned trastuzumab emtansine dose that was actually received, was higher with the 3.6 mg/kg q3w regimen (median 99.7%, range 88%–106%) than with the 2.4 mg/kg qw schedule (median 82%, range 54%–101%). However, since the PK of trastuzumab emtansine is linear at doses ≥ 2.4 mg/kg, an almost 2-fold higher cumulative dose can be

administered within a q3w cycle with a 2.4 mg/kg qw regimen compared with 3.6 mg/kg q3w.<sup>29,30</sup>

Based on a population PK analysis, trastuzumab emtansine has a consistent PK profile with low inter-individual variability (21%–48%) in PK parameters among patients with mBC. Greater baseline tumor burden and lower serum albumin levels, potential indicators of disease severity, resulted in small increases (< 13%) in trastuzumab emtansine clearance (CL). However, trastuzumab emtansine PK was not affected by baseline residual trastuzumab (from prior treatment) or by differences in serum concentrations of HER2 extracellular domain.<sup>35</sup>

An aggregate PK assessment of trastuzumab emtansine was performed with samples from studies TDM3569g, TDM4258g, TDM4374g, and TDM4688g. 36,37 PK parameters for trastuzumab emtansine, total trastuzumab, and DM1 were consistent across the four studies at Cycle 1 and steady state. Trastuzumab emtansine PK was not affected by residual trastuzumab from prior therapy or circulating extracellular domain of HER2. No significant correlations were observed between trastuzumab emtansine exposure and efficacy, thrombocytopenia, or increased concentrations of transaminases. Across the four studies, the incidence of anti-therapeutic antibodies to trastuzumab emtansine was low and detected in 4.5% (13/286) of evaluable patients receiving trastuzumab emtansine q3w.

The PK profile (i.e., maximum concentration [ $C_{max}$ ], area under the serum concentration-time curve [AUC], terminal half-life [ $T_{1/2}$ ], apparent volume of distribution at steady state [ $V_{ss}$ ], and CL) of single-agent trastuzumab emtansine (3.6 mg/kg q3w) is predictable, well characterized, and unaffected by circulating levels of HER2 extracellular domain or residual trastuzumab. Trastuzumab emtansine exposure does not correlate with clinical responses or key AEs. Weekly administration of trastuzumab emtansine in study TDM3568g at a dose of 2.4 mg/kg showed consistent PK data with the q3w dosing schedule.<sup>29</sup>

#### 1.2.2 CAPECITABINE

Capecitabine (Xeloda<sup>®</sup>) is a fluoropyrimidine carbamate with antineoplastic activity. It is an orally administered systemic prodrug of 5'-deoxy-5-fluorouridine (5'-DFUR), which is converted to 5-fluorouracil (5-FU) in the tumor, where it inhibits DNA synthesis and slows down tumor tissue growth. It is approved in combination with docetaxel and as monotherapy in mBC. Please see the national Xeloda<sup>®</sup> prescribing information or Investigator brochure for more information.

The activity of capecitabine as single-agent chemotherapy was initially demonstrated in two multicenter Phase II clinical trials (before testing of HER2 status was standard) in patients with locally advanced or mBC after failure of a taxane and an anthracycline-containing chemotherapy regimen or for whom further anthracycline therapy was not indicated.<sup>38,39</sup> In these trials, a total of 236 patients were treated with capecitabine (1,250 mg/m² bid for 2 weeks followed by 1-week rest period). The ORRs (investigator assessment) were 20% (first trial)

and 25% (second trial). The median TTP was 3.1 months and 3.2 months, respectively. Median OS was 12.6 months and 12.3 months, respectively.

The combination of capecitabine and docetaxel was studied as treatment for locally advanced or mBC after failure of anthracycline-containing chemotherapy in a multicenter randomized controlled Phase III clinical trial (SO14999). In this trial, 255 patients were randomized to treatment with capecitabine (1,250 mg/m² bid for 2 weeks followed by a 1-week rest period) and docetaxel (75 mg/m² as a 1-hour IV infusion q3w) and 256 patients were randomized to treatment with docetaxel alone (100 mg/m² as a 1-hour IV infusion q3w). OS was superior in the capecitabine plus docetaxel combination arm (HR 0.775; p = 0.0126). Median OS was 14.5 months (capecitabine plus docetaxel) *versus* 11.5 months (docetaxel alone). The ORR in the all-randomized population (investigator assessment) was 41.6% (capecitabine plus docetaxel) *versus* 29.7% (docetaxel alone; p = 0.0058). TTP was superior in the capecitabine plus docetaxel combination arm (HR 0.652; p < 0.0001). The median TTP was 6.1 months (capecitabine plus docetaxel) *versus* 4.2 months (docetaxel alone).

This trial led to the randomized Phase II CHAT trial evaluating the addition of capecitabine to first-line trastuzumab and docetaxel for locally advanced or metastatic HER2-positive mBC.<sup>41</sup> PFS was significantly improved with the addition of capecitabine (HR 0.72; median 17.9 months *versus* 12.8 months in patients receiving docetaxel and trastuzumab without capecitabine), although there was no difference in ORR (71% *versus* 73%, respectively).

# 1.2.2.1 Study BO18255: Capecitabine and Trastuzumab in LA/mGC

A global Phase III study (ToGA trial, BO18255) of trastuzumab plus chemotherapy as first-line treatment for advanced HER2-positive GC was conducted in 584 patients previously untreated for HER2-positive inoperable locally advanced or recurrent and/or metastatic adenocarcinoma of the stomach or GEJ. Patients received either capecitabine or fluorouracil combined with cisplatin or the same chemotherapy in combination with trastuzumab. The primary study endpoint was OS, defined as the time from the date of randomization to the date of death from any cause. At the time of the analysis a total of 349 randomized patients had died: 182/290 patients (62.8%) in the control arm and 167/294 patients (56.8%) in the trastuzumab-containing arm. The majority of the deaths were due to events related to the underlying cancer. 18

Most patients enrolled in the study were male (76%); 52.9% were Asian and 37.7% were white. The primary tumor site was the stomach for 81.8% of patients, with the others having GEJ tumors. The addition of trastuzumab to chemotherapy resulted in an increase in median OS from 11.1 months to 13.8 months (HR 0.74, p = 0.0046). ORR (47% *versus* 35%), PFS (median 6.7 *versus* 5.5 months), and TTP (median 7.1 *versus* 5.6 months) were also significantly increased with the addition of trastuzumab to chemotherapy compared with chemotherapy alone.

With regard to OS, a treatment effect could not be excluded in any predefined subgroup, including primary tumor site, histologic subtype, method of determining HER2-positivity, performance status, chemotherapy regimen, age, gender, and region of enrollment. A multivariate analysis for OS showed a consistent result, with an adjusted HR of 0.72 (p = 0.0036); variables found to influence primary outcome included Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1 *versus* 2), prior gastrectomy, and Asian region of enrollment (data on file). A multivariate analysis of OS for patients enrolled in Japan, from which the bulk of Asian patients were enrolled, demonstrated a HR of 0.68. This was consistent with the overall study results.<sup>42</sup>

A pre-planned subgroup analysis by IHC score indicated that positive treatment effects were greater in tumors with higher levels of HER2 expression. Among patients whose tumors had these higher levels of HER2 expression, the median OS was 11.8 months *versus* 16 months (HR = 0.65; 95% CI: 0.51–0.83) and median PFS was 5.5 months *versus* 7.6 months (HR = 0.64; 95 % CI: 0.51–0.79) for chemotherapy *versus* chemotherapy plus trastuzumab respectively. For OS, the HR was 0.75 (95% CI: 0.51–1.11) in the IHC 2+/FISH+ group and 0.58 (95% CI: 0.41–0.81) in the IHC 3+/FISH+ group.<sup>18</sup>

The addition of trastuzumab to chemotherapy did not result in an increased incidence of severe (Grade 3/4) or fatal AEs. There were no additional significant safety issues with trastuzumab used in the treatment of advanced GC over and above those observed when it was used in BC. Taken together, the results of the ToGA trial (BO18255) not only demonstrate the role of HER2 suppression in the treatment of HER2-positive GC but also show that HER2-directed therapies can be added to conventional chemotherapy regimens without substantial increases in side effects.

# 1.2.3 PRECLINICAL DATA OF THE COMBINATION OF TRASTUZUMAB EMTANSINE AND A FLUOROPYRIMIDINE

In preclinical BC models, additive anti-tumor activity was observed with combinations of trastuzumab emtansine and 5-FU (seeFigure 2).<sup>43</sup> In GC models a similar additive effect was observed with trastuzumab emtansine and capecitabine (see Figure 3 [data on file]).

Figure 2 MMTV HER2 Fo5 Mammary Tumor Transplants



T-DM1 = trastuzumab emtansine; 5-FU = 5-fluorouracil

Figure 3 Anti-tumor Activity of Trastuzumab Emtansine in Combination with Capecitabine in NCI-N87

T-DM1 = trastuzumab emtansine; 5-FU = 5-fluorouracil

# 1.3 STUDY RATIONALE AND RISK-BENEFIT ASSESSMENT

# 1.3.1 FOR MBC

At present, mBC remains an incurable disease. The primary goal of treatment is maximizing the patient's survival and quality of life.

HER2-positive breast tumors have been shown to benefit from anti-HER2 therapy. Regimens using the combination of anti-HER2 agents and chemotherapy have demonstrated higher efficacy than single-agent therapy. As a consequence several different combination therapies have been approved for HER2-positive mBC treatment in most countries and are considered the current standard of care.

The combination of capecitabine with anti-HER2 therapies has been shown to be beneficial in patients with HER2-positive mBC. The combination of capecitabine and lapatinib was approved in the United States in March 2007 for the treatment of patients with HER2-positive mBC who have previously received an anthracycline, a taxane, and trastuzumab. In June 2008, the European Commission granted conditional marketing authorization for lapatinib in combination with capecitabine for the treatment of patients with HER2-positive advanced or mBC whose disease has progressed on an anthracycline, a taxane,

and trastuzumab in the metastatic setting. The combination of capecitabine and trastuzumab has demonstrated significant efficacy benefit when compared with capecitabine alone.<sup>9</sup>

The Phase III, TDM4370g trial met its co-primary endpoint of improving PFS (by independent review) and OS compared with the combination of lapatinib and capecitabine (see Section 1.2.1.6).

Based on the studies mentioned above, the combination of trastuzumab emtansine and capecitabine could provide the potential for enhanced anti-tumor efficacy in mBC compared with single-agent trastuzumab emtansine or trastuzumab in combination with chemotherapy. Furthermore, preclinical data suggest that the combination of trastuzumab emtansine and capecitabine has an additive effect (see Section 1.2.3).

Approximately 2,000 patients with BC have been treated in trastuzumab emtansine clinical trials with an acceptable safety profile and a positive risk-benefit ratio. A broad development program is in place to seek approval for indications for mBC. Capecitabine in combination with an anti-HER2 agent is a proven efficacious regimen with a well-established safety profile in mBC. Trastuzumab emtansine and capecitabine have no known significant overlapping toxicities. As part of the Phase I conduct, regular teleconference calls with the investigators will be held to discuss the study treatment risk-benefit profile for each patient. An Independent Data Monitoring Committee (IDMC) will be established with the main responsibility of assessing the risk-benefit for the Phase II part of the study. Therefore, exploring the benefit of combination therapy of trastuzumab emtansine and capecitabine in patients with mBC seems justified.

## 1.3.2 FOR MGC

As for mBC, the primary goal of treatment for metastatic gastric cancer (mGC) is to maximize patients' survival and quality of life.

In HER2-positive gastric tumors, anti-HER2 therapy has shown benefit. In the ToGA study (BO18255), the combination of chemotherapy and trastuzumab significantly improved OS versus chemotherapy alone (see Section 1.2.2.1) in this population. Fluoropyrimidine-based therapies (capecitabine, 5-FU) are the standard of care in mGC in general and were also the most frequent combination agents used in the ToGA trial (BO18255; see Section 1.2.2.1).

Furthermore, preclinical data suggest that the combination of trastuzumab emtansine and capecitabine has an additive effect (see Section 1.2.3).

A development program for trastuzumab emtansine is in place to seek approval for mGC indications. Capecitabine in combination with trastuzumab is a proven efficacious regimen with a well-established safety profile in mGC. Trastuzumab emtansine and capecitabine might have overlapping toxicities and therefore safety monitoring is in place to avoid exposing patients to harm. Therefore,
exploring the benefit of combination therapy of trastuzumab emtansine and capecitabine in patients with mGC seems justified.

In the ToGA study in LA/mGC, trastuzumab exposure was lower than that observed in breast cancer studies. Based on this observation, together with pharmacokinetic results and findings from a Phase I study in mBC, it was considered that a weekly trastuzumab emtansine regimen may provide higher cumulative trastuzumab emtansine exposure than the q3w schedule and was therefore chosen for the Phase I, Cohort 2 part of the present study in LA/mGC. This approach has subsequently been supported by findings from stage I of the adaptive phase II/III BO27952 trial in this setting (see Section 3.3.2.2). In October 2013, the IDMC for the BO27952 trial recommended selection of the weekly 2.4 mg/kg regimen for further evaluation in the phase III part of the trial based on pharmacokinetic, safety, and efficacy data available at the time.

Results from the Phase I part of the study in mGC will be used as supporting information for future studies in the indication.

# 2. OBJECTIVES

# 2.1 PHASE I: MTD-FINDING OF TRASTUZUMAB EMTANSINE AND CAPECITABINE IN MBC

#### 2.1.1 PRIMARY OBJECTIVE

 To determine the MTD of the combination of trastuzumab emtansine and capecitabine in patients with HER2-positive mBC

#### 2.1.2 SECONDARY OBJECTIVES

To assess the:

- PK of trastuzumab emtansine, capecitabine and their metabolites
- Safety of the combination of trastuzumab emtansine and capecitabine
- ORR

# 2.2 RANDOMIZED PHASE II: EXPLORATION OF EFFICACY AND SAFETY IN MBC

#### 2.2.1 PRIMARY OBJECTIVE

To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone in patients with HER2-positive mBC, as measured by ORR by RECIST v.1.1 per investigator local assessment

#### 2.2.2 SECONDARY OBJECTIVES

To assess the safety profile of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone

To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone in patients with HER2-positive mBC, as measured by:

- Time to response (TTR)
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

# 2.3 PHASE I: MTD FINDING OF TRASTUZUMAB EMTANSINE AND CAPECITABINE IN LA/MGC

#### 2.3.1 PRIMARY OBJECTIVE

To determine the MTD of the combination of trastuzumab emtansine and capecitabine in patients with LA/mGC

#### 2.3.2 SECONDARY OBJECTIVES

To assess the:

- PK of trastuzumab emtansine, capecitabine, and their metabolites
- Safety of the combination of trastuzumab emtansine and capecitabine
- ORR

# 3. STUDY DESIGN

# 3.1 DESCRIPTION OF STUDY

This is an international, multicenter Phase I/II dose-finding study of two dosing schedules of trastuzumab emtansine and capecitabine combination therapy in HER2-positive mBC and LA/mGC.

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in Phase I studies in patients with HER2-positive mBC or LA/mGC.

The efficacy and safety of the combination in patients with mBC will also be explored in a randomized, open-label Phase II part of the study.

# 3.1.1 OVERVIEW OF STUDY DESIGN

# **Overview of Study Design**

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with HER2-positive mBC or LA/mGC using a Phase I design, followed by a randomized, open-label Phase II part of the study to explore the efficacy and safety of the combination in patients with HER2-positive mBC. There will be no follow-on randomized exploration of efficacy in mGC. Results from the Phase I study in LA/mGC will be used as supporting information for future studies in the indication.

Cohort 1 for patients with mBC will open first and the MTD will be established. Once the MTD is defined, both the randomized Phase II trial for patients with HER2-positive mBC and the Phase I Cohort 2 for patients with LA/mGC will open.

An overview of the study design is depicted in Figure 4.

# **Duration of Treatment and Patient Follow-up**

<u>Duration of treatment:</u> All patients will be treated until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor. In case of toxicities requiring the discontinuation of capecitabine, single agent trastuzumab emtansine may be continued. In case of toxicities requiring the discontinuation of trastuzumab emtansine, the patient will be followed up until EOS (treatment with capecitabine alone is not allowed).

If at the time of study closure there are patients whose disease has not progressed and who are still receiving study treatment, they will be offered the possibility to continue treatment by enrolling in an extension study at the discretion of the investigator.

<u>Patient follow-up:</u> All patients will be followed up until withdrawal of consent, death, or for up to a maximum of 2 years after the last patient was randomized in the Randomized Phase II part of the study, whichever occurs first.

# **Duration of Study, Database Closure and Data Reporting**

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to last 2 years in total (1 year for the MTD-Finding study in mBC and 1 year for the Phase II Exploration of Efficacy and Safety in mBC). See Section 3.2 for further details about EOS.

Specifically in Phase I, cohort 2, if dose level -2 is too toxic in LA/mGC, recruitment into the LA/mGC cohort will be closed. See Section 3.1.1.3 for details of treatment continuation if patients are still responding to treatment at this time.

Data may be published/presented publicly at the end of each cohort e.g., once the MTD for Cohort 1 for mBC has been defined and the dose for Phase II Exploration of Efficacy and Safety has been selected, and after the prespecified

analyses for the Randomized Phase II exploration of efficacy and safety in mBC. The Clinical Study Report (CSR) will be finalized/published within 1 year after EOS (LPLV).

Figure 4 Overview of Study Design



<sup>&</sup>lt;sup>1</sup> Capecitabine doses are administered daily on Days 1–14 q3w

mBC = metastatic breast cancer; LA/mGC = locally advanced/metastatic gastric cancer; MTD = maximum tolerated dose; q3w = every 3 weeks; qw = weekly.

A schedule of assessments is provided in Appendix 1.

## 3.1.1.1 Overview of Phase I Design in Patients with mBC

An overview of the Phase I study design is depicted in Figure 5.

<sup>&</sup>lt;sup>2</sup> The MTD defined in the mBC Phase I study will be implemented in the mBC Randomized Phase II and mGC Phase I studies

<sup>&</sup>lt;sup>3</sup> Cohort 2 will open to recruit patients with LA/mGC using the MTD defined in Phase I for patients with mBC. Dose Level 1 will not be explored in Cohort 2 (see also Section 3.3.2.2)

<sup>&</sup>lt;sup>4</sup> Stratification factor: Number of prior lines of treatment for metastatic disease (≤1 or >1; excluding single-agent hormones)



Figure 5 Overview of Phase I Dose Finding Study Design

DLT = dose-limiting toxicity: MTD = maximum tolerated dose

#### Determination of the MTD in Patients with mBC

The trial will first investigate the feasibility of the combination of capecitabine and trastuzumab emtansine q3w in one cohort of up to 18 patients, by de-escalating the dose of capecitabine from 750 mg/m² bid to 650 mg/m² bid on Days 1 to 14 q3w with a 3 plus 3 classical Phase I design. Cohort 1 will open first and enroll patients with HER2-positive mBC.

### **Enrollment into Cohort 1**

# MTD-finding in patients with mBC (Phase I)

According to the 3 plus 3 classical study design, Cohort 1 will start with the enrollment of 3 patients at Dose Level 1. Patients will be evaluated for DLTs as specified in the DLT definition (see Section 5.1.4). The dose of trastuzumab emtansine is fixed at 3.6 mg/kg q3w. Three dose levels of capecitabine administered bid on Days 1 to 14 q3w will be tested.

The following doses will be explored in Cohort 1:

<sup>&</sup>lt;sup>1</sup> Repeat with the new dose level until the MTD is established

<sup>&</sup>lt;sup>2</sup> If Dose Level -2 is too toxic (DLT in > 1/6 patients), the study will be terminated.

**Dose Level 1:** 750 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine

**Dose Level -1:** 700 mg/m² capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine

**Dose Level -2:** 650 mg/m<sup>2</sup> capecitabine bid plus 3.6 mg/kg q3w trastuzumab emtansine

The following MTD determining rules will be applied during the MTD-Finding treatment phase:

- Step 1: Three patients will be enrolled at Dose Level 1
- Step 2: The toxicity of Dose Level 1 will be monitored and the following actions taken:
  - a) If none of these 3 patients (0/3) experiences a DLT, the MTD will be established as the current dose level and will need to be confirmed in 3 more patients (to achieve DLTs in ≤ 1/6 patients at that dose level)
  - b) If 1 of the initial 3 patients (1/3) experiences a DLT, an additional 3 patients should be enrolled and treated at the same dose, i.e., Dose Level 1
  - c) If no additional patients experience a DLT (1/6), the MTD will be established as the current dose level
  - d) If 1 or more additional patients experience a DLT (> 1/6), the dose will be de-escalated to the next lowest dose level. If no more than 1 patient experiences a DLT (≤ 1/6) after dose de-escalation, the dose will be considered the MTD and, following IDMC recommendation, will be further explored in the Randomized Phase II part of the study. Dose re-escalation will not be allowed. If 2 or more patients experience a DLT (> 1/6) after dose de-escalation, de-escalation should continue to the next lowest dose level. Based on the DLT findings, the next dose level may be considered the MTD and, following IDMC recommendation, be further explored in the Randomized Phase II part of the study or the study may be terminated if DLTs occur in > 1/6 patients at Dose Level -2.

In order to define the dose for the Randomized Phase II Exploration of Efficacy and Safety part of the study, evaluation will include not only the DLTs during Cycle 1 but also all available safety information during the subsequent cycles. The dose level considered optimal will be the dose level selected to proceed to the Phase II and LA/mGC parts of the study.

Once the appropriate dose of study medication is established, the Randomized Phase II part of the study and Phase I, Cohort 2 will open as shown in Figure 4.

# 3.1.1.2 Overview of Phase II: Exploration of Efficacy and Safety in Patients with mBC

After review of safety data from Part 1, cohort 1, the IDMC recommended a regimen of capecitabine 700 mg/m² bid days 1–14 in combination with trastuzumab emtansine 3.6 mg/kg q3w for further evaluation. The Phase II part of the study will explore the efficacy and safety of this recommended regimen compared with trastuzumab emtansine alone in patients with HER2-positive mBC. See Section 3.1.1 for details of duration of treatment.

Approximately 160 additional patients with HER2-positive mBC will be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to the Phase II part of the study; however, they will be followed-up until end of study (EOS).

# 3.1.1.3 Overview of Phase I Design in LA/mGC Patients

#### Determination of the MTD in Patients with LA/mGC

Cohort 2 will enroll patients with HER2-positive LA/mGC. Trastuzumab emtansine will be administered qw at a fixed dose of 2.4 mg/kg and capecitabine will be started at 700 mg/m² bid, the MTD defined for patients with mBC in Cohort 1.

### **Enrollment into Cohort 2**

Cohort 2 will open with a 3 plus 3 classical design to investigate the feasibility of combination therapy of capecitabine and trastuzumab emtansine in up to 12 patients with LA/mGC. The capecitabine dose will be de-escalated from the starting dose of 700 mg/m² bid (the MTD recommended in Cohort 1).

The dose levels for de-escalation of capecitabine will be the same as described for Cohort 1, except for Dose Level 1, which will not be explored in patients with mGC (see also Section 3.3.2.2).

If Dose Level -1 (700 mg/m<sup>2</sup> bid, the MTD recommended in cohort 1) is well tolerated (DLT in  $\leq$  1/6), this dose will be established as the MTD for LA/mGC.

- If Dose Level -1 is not tolerated in Cohort 2 (DLT in > 1/3 or > 1/6 patients), de-escalation will be to Dose Level -2.
- If Dose Level -2 is not tolerated in Cohort 2 (DLT in > 1/6), the combination will be considered not feasible in LA/mGC and Cohort 2 will be terminated. Patients who, at that time, experience response according to RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the Steering Committee (SC).

#### 3.1.1.4 Number of Patients

Overall, it is anticipated that the maximum number of patients enrolled into the study will be approximately 190.

# Phase I, Cohort 1: mBC

Between 6 and 18 patients will be enrolled into Cohort 1 to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with mBC.

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

For this part of the study, a total of approximately 160 patients with mBC will be randomized.

### Phase I, Cohort 2: mGC

After the MTD in Cohort 1 has been established, 3–12 patients will be enrolled into Cohort 2 to determine the MTD of capecitabine in combination with trastuzumab emtansine in patients with mGC.

#### 3.1.1.5 Number of Centers

This is a multicenter, international study.

# 3.1.2 STEERING COMMITTEE

A SC has been established for this study. Initially, it is composed of the investigators participating in the Phase I, Cohort 1 part of the study and one medical representative and one statistician of the Sponsor. The study design and DLT definition have been developed by the SC. See the SC Charter for further information

The SC will collectively review the status of the ongoing patients in Phase I on a regular basis. The SC will adjudicate in the event of DLTs that are not covered by the existing DLT criteria.

# 3.1.3 INDEPENDENT DATA MONITORING COMMITTEE

An IDMC will review the safety outcomes for patients enrolled in Phase I, Cohort 1 and recommend whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 25, 75, and 150 patients have received at least 3 cycles (Cycle 3 Day 21) of treatment in the Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II part of the study or as requested.

# 3.2 END OF STUDY

EOS is defined as the last patient last visit (LPLV) at the end of the follow-up period, as defined in Section 3.1.1. This will be the last data collection point,

which can be a clinic visit or a laboratory sample. LPLV is expected to occur approximately 2 years after the last patient has been randomized into the Phase II part of the trial.

# 3.3 RATIONALE FOR STUDY DESIGN

# 3.3.1 RATIONALE FOR PATIENT GROUP SELECTION

Nonclinical studies indicate that the sensitivity of cancer cells to trastuzumab emtansine requires HER2 overexpression, and measurement of such expression is a standard of care in determining eligibility for trastuzumab therapy (see the Herceptin® national prescribing information). Measurement of HER2 gene amplification has traditionally been performed using IHC. HER2 gene amplification determined by ISH has also proven to be a reliable method for demonstrating HER2-positive status.<sup>44</sup>

This study will enroll patients diagnosed with HER2-positive mBC or LA/mGC. Capecitabine is an established chemotherapy for both diseases. In patients with HER2-positive mBC or LA/mGC, anti-HER2 therapy has demonstrated activity. Furthermore, the combination of anti-HER2 therapy and capecitabine has been shown to be efficacious in both mBC<sup>9,10</sup> and LA/mGC.<sup>18</sup> Eligible patients for this study will have incurable mBC or LA/mGC overexpressing HER2.

#### 3.3.1.1 Rationale for Phase I

The 3 plus 3 design is a well-established and well-known method for Phase I studies. PK parameters will be collected and analyzed to investigate the PK interaction of the drugs under investigation.

The capecitabine dose evaluated in combination with trastuzumab and docetaxel in the CHAT trial was 950 mg/m² bid. However, retrospective evaluations and post hoc analyses of early dose reduction suggest that lower starting doses of capecitabine offer similar efficacy with better tolerability. Therefore the capecitabine starting dose selected in combination with trastuzumab emtansine for the MTD-Finding Phase I part of the present study was 750 mg/m² bid, taking into account the aim of maintaining the good tolerability of trastuzumab emtansine while benefitting from synergy observed between the two agents in nonclinical studies.

The combination of T-DM1 and capecitabine was evaluated with a de-escalation study design. Following the emergence of two DLTs (grade 3 vomiting, grade 3 elevated AST/ALT) at the starting dose of 750 mg/m² bid (days 1–14 q3w) in combination with trastuzumab emtansine 3.6 mg/kg q3w, a de-escalated dose cohort was opened to evaluate capecitabine 700 mg/m² bid combined with the same dose of trastuzumab emtansine. At this dose no DLTs were observed in the six patients treated, and of note, none of the patients had experienced grade ≥3 AEs in cycles delivered after the DLT evaluation period.<sup>45</sup> Following review of safety data from patients treated at these two dose levels, the IDMC

recommended the regimen of capecitabine 700 mg/m² bid combined with trastuzumab emtansine 3.6 mg/kg q3w for the phase II exploration of efficacy and safety.

In the ToGA study in LA/mGC, trastuzumab exposure was lower than that observed in breast cancer studies. A weekly trastuzumab emtansine regimen may provide higher cumulative trastuzumab emtansine exposure than the q3w schedule and was therefore chosen for the Phase I, Cohort 2 part of the present study in LA/mGC. This approach has subsequently been supported by findings from stage I of the adaptive phase II/III BO27952 trial in this setting (see Section 3.3.2.2).

# 3.3.1.2 Rationale for Randomized Phase II

The Randomized Phase II part of the study is designed to explore the efficacy and safety of the combination recommended following the Phase I MTD-Finding phase (trastuzumab emtansine 3.6 mg/kg in combination with capecitabine 700 mg/m²) compared with trastuzumab emtansine alone.

# 3.3.2 RATIONALE FOR INVESTIGATIONAL MEDICINAL DOSE SELECTION

#### 3.3.2.1 In Patients with mBC

In study TDM3569g, the MTD of trastuzumab emtansine administered by IV infusion q3w was 3.6 mg/kg. As described in Section 1.2, clinical activity has been observed at a dose of 3.6 mg/kg q3w in two Phase II studies of single-agent trastuzumab emtansine in patients with heavily pre-treated HER2-positive mBC (protocol TDM4258g³¹ and protocol TDM4374g³²), in patients who had not received prior chemotherapy for metastatic disease (TDM4450g²6), and subsequently in the randomized phase III trials.²7,28

Capecitabine doses have been selected as being in the range of efficacious doses for single-agent or combination use. The doses selected are within the dosing range included in the Xeloda® Summary of Product Characteristics (SmPC) and therefore are considered to be efficacious.

#### 3.3.2.2 In Patients with mGC

In the ToGA study (BO18255) evaluating trastuzumab in combination with chemotherapy for mGC, patients with higher drug exposure had a greater benefit than those with lower exposure.<sup>46</sup> As a consequence, an ongoing randomized, open-label, multicenter Phase IIIb study is comparing two trastuzumab dosing regimens, each in combination with cisplatin/capecitabine chemotherapy, as first-line therapy in patients with HER2-positive metastatic gastric or GEJ adenocarcinoma (Study BO27798).

In TDM3569g (see Section 1.2.1.1), the qw administration of 2.4 mg/kg of trastuzumab emtansine resulted in higher exposure than q3w dosing (see

Section 1.2.1.8).<sup>29,30</sup> Therefore, this dose may result in larger clinical benefit for patients with mGC.

In the ongoing randomized adaptive phase II/III BO27952 trial evaluating trastuzumab emtansine versus the investigator's choice of taxane therapy in unrectable LA/mGC, two trastuzumab emtansine regimens were evaluated in stage I: 3.6 mg/kg q3w and 2.4 mg/kg qw. In October 2013, the IDMC for the BO27952 trial recommended selection of the weekly 2.4 mg/kg regimen for further evaluation in the phase III part of the trial based on pharmacokinetic, safety, and efficacy data available at the time. This recommendation provides further support for using the weekly regimen in Phase I, Cohort 2 of the present trial.

In Cohort 2, the starting dose of capecitabine will be 700 mg/m² bid (the MTD from Cohort 1 in mBC) in order to minimize the exposure of patients to suboptimal treatment. The dose of capecitabine can be de-escalated if needed.

#### 3.3.2.3 Rationale for Duration of Treatment

Treatment will be given until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor (see Section 3.1.1 for full information). As of 1 January 2010, of 237 patients enrolled in studies TDM3569g, TDM4258g, and TDM4374g receiving trastuzumab emtansine at 3.6 mg/kg, approximately 30% have tolerated more than 12 cycles, with 14.8% having received more than 17 cycles. Twenty patients (8.4%) have discontinued trastuzumab emtansine due to AEs and 24 patients (10.1%) required dose reductions in trastuzumab emtansine because of AEs. In the absence of unacceptable toxicity, patients with mBC are generally treated until PD. Further support for treatment until PD comes from the EMILIA randomized phase III trial.<sup>27</sup> Among the 490 patients randomized to trastuzumab-emtansine, only 29 (5.9%) discontinued because of adverse events.

Capecitabine will be given until PD, in accordance with Xeloda<sup>®</sup> national prescribing information.

# 3.3.3 PHARMACOKINETIC SAMPLING RATIONALE

PK is studied only in the Phase I (MTD-Finding) parts (both cohorts 1 and 2). The PK sampling rationale is to characterize the PK of trastuzumab emtansine and capecitabine and their metabolites, to assess any potential drug-drug interaction when trastuzumab emtansine is given in combination with capecitabine, and to explore potential correlations between drug exposure and measures of both efficacy (ORR) and toxicity (alanine transaminase [ALT]/AST, platelets, etc.), if data allow.

# 3.4 OUTCOME MEASURES

# 3.4.1 PHASE I: MBC

# 3.4.1.1 Primary Outcome Measure

The main objective for Phase I is to determine the MTD of capecitabine when combined with trastuzumab emtansine.

# 3.4.1.2 Secondary Outcome Measure

The secondary outcome is ORR, based on best overall response (BOR) rate according to RECIST v.1.1, per investigator local assessment.

# 3.4.1.3 Primary Safety Outcome Measure

The primary safety outcome measure is to establish the MTD. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination and will be summarized for each treatment dosage.

# 3.4.1.4 Secondary Safety Outcome Measures

Safety endpoints will be summarized for each treatment dosage:

- Incidence, nature, and severity of AEs, according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v. 4.0
- Incidence, nature, and severity of SAEs, according to NCI CTCAE v. 4.0
- Incidence and nature of Grade ≥3 AEs
- Incidence, nature, and severity of AEs of special interest (AESIs), according to NCI CTCAE v. 4.0
- Fatal AEs and their causes
- Laboratory parameters
- LVEF
- Exposure to study medication
- Physical examination
- ECOG performance status
- Premature withdrawal from study medication and/or study

## 3.4.1.5 Pharmacokinetic Outcome Measures

The PK outcome measures to be assessed in patients receiving trastuzumab emtansine and capecitabine will include:

 Serum concentrations of trastuzumab emtansine (conjugated drug) and total trastuzumab (free and conjugated to DM1)

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 4, 23 Mar 2016

- Plasma concentration of DM1
- Plasma concentration of capecitabine and its active metabolite 5-FU
- Total exposure (e.g., AUC)
- C<sub>max</sub>
- CL
- V<sub>d</sub>
- T<sub>1/2</sub>

# 3.4.2 RANDOMIZED PHASE II: EXPLORATION OF EFFICACY AND SAFETY IN MBC

The primary and secondary efficacy outcome measures will be presented for each treatment group.

# 3.4.2.1 Primary Efficacy Outcome Measure

The primary outcome measure is ORR by investigator assessment, based on BOR (defined as the best response recorded from randomization into the Phase II part of the study and until PD, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first) according to RECIST v.1.1 (See <u>Appendix 3</u>).

# 3.4.2.2 Secondary Efficacy Outcome Measures

Secondary efficacy outcomes include:

- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

# 3.4.2.3 Primary Safety Outcome Measure

A primary safety outcome is defined only for Phase I.

# 3.4.2.4 Secondary Safety Outcome Measures

The summary of safety endpoints will be presented for each treatment group:

- Incidence, nature, and severity of AEs, according to NCI CTCAE v. 4.0
- Incidence, nature, and severity of SAEs, according to NCI CTCAE v. 4.0

- Incidence and nature of Grade ≥3 AEs
- Incidence, nature, and severity of AESIs, according to NCI CTCAE v. 4.0
- Fatal AEs and their causes
- Events to monitor
- Laboratory parameters
- LVEF
- Exposure to study medication
- Physical examination
- ECOG performance status
- Premature withdrawal from study medication and/or study

#### 3.4.2.5 Pharmacokinetic Outcome Measures

Not applicable for Phase II.

## 3.4.3 Phase I: LA/MGC

# 3.4.3.1 Primary Outcome Measure

The main objective for Phase I is to determine the MTD of capecitabine when combined with trastuzumab emtansine. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination and will be summarized for each treatment dosage.

# 3.4.3.2 Secondary Efficacy Outcome Measure

The secondary (efficacy) outcome is ORR, based on BOR rate according to RECIST v.1.1 according to investigator assessment.

# 3.4.3.3 Secondary Safety Outcome Measures

Safety endpoints will be summarized for each treatment dosage:

- Incidence, nature, and severity of AEs, according to NCI CTCAE v. 4.0
- Incidence, nature, and severity of SAEs, according to NCI CTCAE v. 4.0
- Incidence and nature of Grade ≥3 AEs
- Incidence, nature, and severity of AESIs, according to NCI CTCAE v. 4.0
- Fatal AEs and their causes
- Events to monitor
- Laboratory parameters
- LVEF

#### Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 4, 23 Mar 2016

- Exposure to study medication
- Physical examination
- ECOG performance status
- Premature withdrawal from study medication and/or study

#### 3.4.3.4 Pharmacokinetic Outcome Measures

The PK outcome measures to be assessed in patients receiving trastuzumab emtansine and capecitabine will include:

- Serum concentrations of trastuzumab emtansine (conjugated drug) and total trastuzumab (free and conjugated to DM1)
- Plasma concentration of DM1
- Plasma concentration of capecitabine and its active metabolite 5-FU
- Total exposure (e.g., AUC)
- Cmax
- CL
- V<sub>d</sub>
- T<sub>1/2</sub>

# 4. MATERIALS AND METHODS

# 4.1 PATIENTS

# 4.1.1 PATIENTS WITH MBC

This study will enroll patients with HER2-positive BC with histologically or cytologically confirmed metastatic disease that is amenable to combination treatment with trastuzumab emtansine and capecitabine.

Patients with mBC must have received at least one prior treatment regimen for early or metastatic disease, which included a chemotherapy agent and trastuzumab either separately or in combination. In both study parts (Phase I and II), only patients whose HER2 tumor status was locally scored as IHC 3+ or in situ hybridization (ISH) positive will be eligible.

# 4.1.2 LA/MGC PATIENTS

This study will enroll patients with HER2-positive GC with histologically or cytologically confirmed inoperable LA/mGC that is amenable to combination treatment with trastuzumab emtansine and capecitabine.

Patients with mGC must not have received prior chemotherapy for advanced/metastatic disease, and only patients with HER2-positive primary

tumor or metastasis as assessed by the central laboratory will be allowed to enroll in the mGC part of the study.

### 4.1.3 INCLUSION CRITERIA

#### 4.1.3.1 For Patients with mBC

Patients must meet the following criteria for study entry:

- 1. Male or female
- 2. Age ≥ 18 years old
- 3. Signed informed consent before any study-specific procedure
- 4. Able and willing to comply with the protocol
- 5. Negative serum pregnancy test for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in the medical history confirming that the patient is not of childbearing potential.
- 6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 7 months after the last dose of study treatment (see Section 5.2.4).
- 7. ECOG performance status of 0, 1, or 2
- 8. Blood:
  - a) Platelet count > 100,000 cells/mm<sup>3</sup>
  - b) International normalized ratio (INR) < 1.5
  - c) Absolute neutrophil count (ANC) > 1,500 cells/mm<sup>3</sup>
  - d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.
- 9. Liver function:
  - a) Total bilirubin ≤ 1.5 × upper limit of normal (ULN) or direct bilirubin ≤1.5
    × ULN in patients with documented Gilbert's syndrome.
  - b) Serum glutamic oxaloacetic transaminase (SGOT)/AST and serum glutamic pyruvic transaminase (SGPT)/ALT ≤ 2.5 × ULN
  - c) Alkaline phosphatase  $\leq 2.5 \times ULN$ . In patients with bone metastases: alkaline phosphatase  $\leq 5 \times ULN$
  - d) Evidence of stable liver function during the month prior to enrollment with liver function test (LFT) fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin).

#### 10. Renal function:

 a) Serum creatinine of < 177 μmol/L or calculated creatinine CL > 50 mL/min. If urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate ≤ 1 g of protein/24 hours

#### 11. Cardiac function:

- a) LVEF ≥ 50% by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan
- 12. Life expectancy ≥ 2 weeks
- 13. Histologically or cytologically confirmed BC
- 14. HER2-positive disease, defined as IHC 3+ or ISH positive
- 15. Tumor block or 8 slides available for retrospective central confirmation of HER2-positivity (central confirmation not necessary for enrollment).
- 16. mBC with at least one measurable lesion according to RECIST v.1.1
- 17. Disease progression on at least one prior regimen containing trastuzumab and chemotherapy either separately or in combination. Patients may be eligible to receive study therapy in the first-line setting if trastuzumab and chemotherapy were given in the [neo]adjuvant setting.
- 18. Patients must have recovered from previous treatments

#### 4.1.3.2 For Patients with LA/mGC

Patients must meet the following criteria for study entry:

- Male or female
- 2. Age ≥ 18 years old
- 3. Signed informed consent before any study-specific procedure
- 4. Able and willing to comply with the protocol
- 5. Negative serum pregnancy test for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 12 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in the medical history confirming that the patient is not of childbearing potential
- 6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 7 months after the last dose of study treatment (see Section 5.2.4)
- 7. ECOG performance status of 0, 1, or 2

#### 8. Blood:

- a) Platelet count > 100,000 cells/mm<sup>3</sup>
- b) INR < 1.5
- c) ANC  $> 1,500 \text{ cells/mm}^3$
- d) Hemoglobin > 9.0 g/dL. Patients are allowed to have received transfusion to achieve this level.

# 9. Liver function:

- a) Total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤1.5 × ULN in patients with documented Gilbert's syndrome
- b) SGOT/AST and SGPT/ALT ≤ 2.5 × ULN
- c) Alkaline phosphatase ≤ 2.5 × ULN. In patients with bone metastases: alkaline phosphatase ≤ 5 × ULN
- d) Evidence of stable liver function in the month prior to enrollment with LFT fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin).

#### 10. Renal function:

 a) Serum creatinine of < 177 μmol/L or calculated creatinine CL > 50 mL/min. If urine dipstick for proteinuria is ≥ 2+ at baseline, the patient must undergo 24-hour urine collection and demonstrate ≤ 1 g of protein/24 hours

# 11. Cardiac function:

- a) LVEF ≥ 50% by ECHO or MUGA scan
- 12. Life expectancy ≥ 2 weeks
- 13. Histologically or cytologically confirmed mGC or locally advanced GC
- 14. HER2-positive tumor (primary tumor or metastatic lesion), defined as either IHC 3+ or IHC 2+ and ISH+, prospectively confirmed by a Sponsor-designated central laboratory prior to enrollment. ISH positivity is defined as a ratio of ≥ 2.0 for the number of HER2 gene copies to the number of signals for CEP17.
  - a) Archival tumor samples obtained from primary or metastatic sites are acceptable.
  - b) Invasive tumor for central confirmation of HER2 status is required.
  - c) A formalin-fixed paraffin-embedded (FFPE) tissue block with at least 5 mm of invasive tumor for central confirmation is preferred. If FFPE tissue blocks (or partial block) are unavailable due to country or site regulations, a minimum of 8 freshly cut unstained slides MUST be available for central review of HER2 status.

#### 15. Inoperable LA/mGC

# 4.1.4 EXCLUSION CRITERIA

#### 4.1.4.1 For Patients with mBC

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half-lives, whichever is longer
  - b) Hormonal therapy within 14 days
  - c) Trastuzumab within 21 days
- 2. Prior treatment with trastuzumab emtansine or prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine
- 3. Prior treatment with capecitabine
- 4. History of severe and unexpected reactions to fluoropyrimidine or known hypersensitivity to fluorouracil
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogues, such as brivudine
  - b) Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
  - c) Known complete absence of DPD activity.
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m<sup>2</sup>
  - b) Epirubicin > 900 mg/m<sup>2</sup>
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m<sup>2</sup>
- 8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 28 days before first study drug administration
- 9. Current peripheral neuropathy of Grade ≥ 3 according to NCI CTCAE, v. 4.0
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above.
- 11. Current unstable ventricular arrhythmia requiring treatment

- 12. History of symptomatic CHF (New York Heart Association [NYHA] Classes II–IV)
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
- 15. Severe dyspnea at rest due to complications of advanced malignancy or currently requiring continuous oxygen therapy
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation
- 20. Current known active infection with human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C virus (HBV/HCV)
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Lapatinib ≤ 14 days before first study drug administration
- 22. Previous radiotherapy for the treatment of mBC is not allowed if:
  - a) The last fraction of radiotherapy has been administered within 14 days prior to first study drug administration (28 days for patients with radiotherapy to control symptoms of brain metastases, see exclusion criterion 8).
  - b) More than 25% of marrow-bearing bone has been irradiated.
  - c) Any acute toxicity has not resolved to Grade ≤ 1 before first study drug administration.

#### 4.1.4.2 For Patients with LA/mGC

- 1. Prior treatments before first study treatment:
  - a) Investigational therapy within ≤ 28 days or 5 half-lives, whichever is longer
  - b) Hormonal therapy within 14 days
  - c) Trastuzumab within 21 days
- 2. Prior treatment with trastuzumab emtansine or prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received prior trastuzumab emtansine

- 3. Prior treatment with capecitabine
- 4. History of severe or unexpected reactions to fluoropyrimidine or known hypersensitivity to fluorouracil
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogs, such as brivudine
  - b) Rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
  - c) Known complete absence of DPD activity.
- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 500 mg/m²
  - b) Epirubicin > 900 mg/m<sup>2</sup>
  - c) Mitoxantrone > 120 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m² doxorubicin.
- Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control symptoms within 28 days before first study drug administration
- 9. Current peripheral neuropathy of Grade ≥ 3 according to NCI CTCAE, v. 4.0
- 10. History of other malignancy within the last 5 years, except for appropriately treated carcinoma *in situ* of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above
- 11. Current unstable ventricular arrhythmia requiring treatment
- 12. History of symptomatic CHF (NYHA Classes II-IV)
- 13. History of myocardial infarction or unstable angina within 6 months prior to first study drug administration
- 14. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
- 15. Severe dyspnea at rest due to complications of advanced malignancy or currently requiring continuous oxygen therapy
- 16. Clinically significant malabsorption syndrome or inability to take oral medication
- 17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)

- 18. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
- 19. Current pregnancy or lactation
- 20. Current known active infection with HIV, HBV, and/or HCV
  - a) For patients who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
- 21. Previous chemotherapy for advanced/metastatic disease
  - a) Prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrollment into the study
- 22. Lapatinib ≤ 14 days before first study drug administration

# 4.1.5 PATIENT REPLACEMENT POLICY

None of the patients in the Phase I part of the study may be replaced unless approved by the entire SC. Phase II patients will not be replaced.

# 4.2 METHOD OF TREATMENT ASSIGNMENT

In the Randomized Phase II part of the study, patients will be randomized to receive either the combination of trastuzumab emtansine and capecitabine or trastuzumab emtansine alone. Patients are stratified according to the number of prior lines of treatment for metastatic disease (≤ or > , excluding single-agent therapy).

This is an open-label randomized study; therefore, no blinding will be used.

#### 4.3 STUDY TREATMENT

# 4.3.1 FORMULATION, PACKAGING, AND HANDLING

# 4.3.1.1 Trastuzumab Emtansine

Trastuzumab emtansine is provided as a single-use, lyophilized formulation in a colorless 20 mL Type I glass vial containing 160 mg of trastuzumab emtansine, closed by means of a FluroTec coated stopper and an overseal with flip-off cap. Upon receipt of trastuzumab emtansine, vials should be refrigerated at 2–8°C (36–46°F) until use. THE VIAL MUST NOT BE FROZEN OR SHAKEN. Trastuzumab emtansine must be stored in the original carton to protect it from light. Do not use the product beyond the expiration date provided by the manufacturer. Any remaining medication should be discarded.

All vials of trastuzumab emtansine should be handled by appropriately trained site staff wearing gloves and using appropriate procedures in place at the clinical

site for preparation of chemotherapeutic drugs. Vials should be visually inspected upon receipt to ensure that they are intact without exterior contamination. Discard any cracked vials and report vials with surface contamination to the clinical site manager for assessment.

The lyophilized product should be reconstituted using sterile water for injection (SWFI). Using a new syringe, 8 mL SWFI should be added to the vial and the vial swirled gently until the product is completely dissolved. The vial should not be shaken. The resulting product contains 20 mg/mL trastuzumab emtansine, 10 mM sodium succinate, pH 5.0, 60 mg/mL sucrose, and 0.02% (w/v) polysorbate 20. Each 20 mL vial contains enough trastuzumab emtansine to allow delivery of 160 mg trastuzumab emtansine. The reconstituted product contains no preservative and is intended for single use only.

The vial should be inspected to ensure the reconstituted product is a clear colorless solution, and is free of particulates before proceeding. Drug from any vial that appears abnormal upon inspection should not be administered to patients. Using a new syringe, the indicated volume of trastuzumab emtansine solution should be removed from the vial(s) and added to the IV bag containing at least 250 mL of 0.45% sodium chloride (preferred) or 0.9% sodium chloride injection and gently inverted to mix the solution. A 0.22 micron non-protein adsorptive polyethersulfone in line filter is recommended when using 0.45% sodium chloride and required when using 0.9% sodium chloride injection. The solution of trastuzumab emtansine should not be shaken.

The solution of trastuzumab emtansine for infusion should be used immediately. If not used immediately, storage times should not be longer than 24 hours at 2–8°C (36–46°F) for solutions of trastuzumab emtansine diluted in polyvinyl chloride (PVC) or latex free PVC-free polyolefin, polypropylene, or polyethylene bags containing 0.45% or 0.9% Sodium Chloride for Injection.

For additional details, please refer to the current version of the trastuzumab emtansine Investigator's Brochure.

# 4.3.1.2 Capecitabine

The following information has been obtained from the Xeloda® European Union (EU) SmPC and US Xeloda® Package Insert.

Capecitabine is available as biconvex, oblong, film-coated tablets, available as follows:

- 150 mg tablets: color, light peach; engraving, XELODA on one side, 150 on the other; packs of 60
- 500 mg tablets: color, peach; engraving, XELODA on one side, 500 on the other; packs of 120

Capecitabine tablets should not be stored above 30°C.

#### 4.3.2 DOSAGE AND ADMINISTRATION

#### 4.3.2.1 For Patients with mBC

#### **Trastuzumab Emtansine**

Trastuzumab emtansine will be administered on Day 1 q3w at a dose of 3.6 mg/kg IV (see Appendix 1). The total dose will be calculated based on the patient's weight on Day 1 of each cycle (or up to 3 days before) with no upper limit.

If the timing of trastuzumab emtansine coincides with a holiday that precludes the procedure, the procedure should be performed within 3 business days of the scheduled date and, when possible, on the earliest following date, with subsequent protocol-specified procedures rescheduled accordingly.

The first infusion of trastuzumab emtansine will be administered over 90 minutes (±10 minutes). Infusions may be slowed or interrupted for patients experiencing infusion-associated symptoms. Vital signs must be assessed before and after dose administration. Following the initial dose, patients will be observed for at least 90 minutes for fever, chills, or other infusion-associated symptoms. If prior infusions were well tolerated (without any signs or symptoms of infusion reactions), subsequent doses of trastuzumab emtansine may be administered over 30 minutes (±10 minutes), with a minimum 30-minute observation period following infusion. Local health authority guidelines must be followed with regard to further observation and monitoring, if applicable.

Pre-medication for nausea and infusion reactions (e.g., acetaminophen or other analgesics, antihistamines such as diphenhydramine, or corticosteroids) may be given at the investigator's discretion.

# Capecitabine

Capecitabine will be administered twice a day, orally for 14 days followed by a 7-day rest period at the Dose Levels described in Section 3.1.1. Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Capecitabine doses can be delayed for up to 4 hours, while keeping the minimal interval of 8 hours between the doses.

Rounding of the dose, based on 150 and 500 mg strength tablets, will be allowed to the nearest dose per patient body surface area (BSA).

If a dose is missed, the patient should skip that dose. The patient should not double the dose during the next administration.

Guidelines for dosage modification and treatment interruption or discontinuation are provided in Section 5.1.

#### 4.3.2.2 For Patients with LA/mGC

#### **Trastuzumab Emtansine**

Trastuzumab emtansine will be administered on Day 1 qw at a dose of 2.4 mg/kg IV (see Appendix 1). The total dose will be calculated based on the patient's weight on Day 1 of each cycle (or up to 3 days before) with no upper limit.

Administration time and observation period are described in Section 4.3.2.1 for trastuzumab emtansine.

Guidelines regarding timing delays and infusion times are the same as for patients with mBC, as is the accepted pre-medication.

# Capecitabine

Capecitabine will be administered at a starting dose of 700 mg/m² bid, orally, for 14 days followed by a 7-day rest period (the dose level determined as the MTD in cohort 1, with de-escalation as described in section 3.1.1.3. Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Capecitabine doses can be delayed for up to 4 hours, while keeping the minimal interval of 8 hours between the doses.

If a dose is missed, the patient should skip that dose. The patient should not double the dose at the next administration.

Guidelines for dosage modification and treatment interruption or discontinuation are provided in Section 5.1.

### 4.3.3 INVESTIGATIONAL MEDICINAL PRODUCT ACCOUNTABILITY

All investigational medicinal products (IMPs) required for completion of this study (trastuzumab emtansine and capecitabine) will be provided by the Sponsor. The investigational site will acknowledge receipt of IMPs, using the interactive voice/web recognition system (IxRS) to confirm the shipment condition and content. Any damaged shipments will be replaced.

IMPs will be either disposed of at the study site according to the study site's institutional standard operating procedure or returned to the Sponsor with the appropriate documentation. The site's method of IMP destruction must be agreed upon by the Sponsor. The site must obtain written authorization from the Sponsor before any IMP is destroyed, and IMP destruction must be documented on the appropriate form.

Accurate records of all IMPs received at, dispensed from, returned to, and disposed of by the study site should be recorded on the Drug Inventory Log.

# 4.3.4 Post-trial Access to Extension Study

Post-trial access to trastuzumab emtansine and capecitabine will be performed as described in Section 3.1.1, Duration of Treatment and Patient Follow-Up. If a

patient decides to withdraw from the study, no post-trial access will be granted. Currently, the Sponsor does not have any plans to provide other study interventions to patients after conclusion of the study or any earlier patient withdrawal

# 4.4 CONCOMITANT AND EXCLUDED THERAPIES

#### 4.4.1 PERMITTED THERAPY

Concomitant therapy and pre-medication are defined as non-IMPs.

Concomitant therapy includes any prescription medication, over-the-counter preparation, or herbal therapy between the 14 days preceding first treatment and the Study Treatment Discontinuation Visit. Afterwards, only anti-cancer therapies will be collected as part of the survival follow-up.

Pre-medication is allowed according to standard practice guidelines.

No pre-medication for the first infusion of trastuzumab emtansine is required; however, pre-medication is allowed at the investigator's discretion.

Concomitant use of erythropoiesis-stimulating agents is allowed if clinically indicated in accordance with local prescribing guidelines.

Palliative radiotherapy is permitted to treat pre-existing painful bone metastases or to treat brain metastases (for patients who have disease control outside of the brain). Please contact the Medical Monitor for approval. If the Medical Monitor cannot be reached because of time zone differences, radiotherapy may be administered, but the Medical Monitor should still be informed.

Other medications considered necessary for the patient's safety and well-being may be given at the discretion of the investigator. Use of bisphosphonates or denosumab is permitted for the control of bone pain, prevention and/or treatment of bony metastases, and treatment of osteoporosis. If bisphosphonates are required for the treatment of symptomatic malignancy-associated hypercalcemia, tumor assessments should be performed to assess for potential PD.

## 4.4.2 PROHIBITED THERAPY

During the study, use of the therapies described below is prohibited until discontinuation of study treatment (collectively, these will be referred to as non-protocol therapy).

Any therapies intended for the treatment of cancer, other than trastuzumab emtansine, whether they are approved by national health authorities or experimental, including cytotoxic chemotherapy, immunotherapy, hormonal therapy (other than megestrol acetate), and biologic or targeted agents (other than granulocyte colony-stimulating factor and erythropoiesis-stimulating agents), are prohibited.

Radiotherapy for unequivocal PD is not permitted while on study treatment, with the exception of new brain metastases or isolated progression of previously treated brain lesions. Patients who have disease control outside of the brain, defined as continued PR or CR of any duration, or SD for ≥ 3 months, but who have developed brain metastases that are treatable with radiation will be allowed to continue to receive study therapy until they either experience systemic progression of their disease and/or further progression in the brain that cannot be treated with additional radiation. Patients must not miss more than one cycle of study treatment for the treatment of their brain metastases and must have an ECOG performance status of 0, 1, or 2 to continue on therapy. The Medical Monitor should be informed before a decision is made to resume study treatment after radiotherapy for brain metastases.

## 4.5 STUDY ASSESSMENTS

All patients will be closely monitored for safety and tolerability during all cycles of therapy and at the safety follow-up visit:

- Visits will be based on a q3w cycle for mBC
- Visits will be based on a qw cycle for mGC

Study assessments are outlined in this section and in Appendix 1.

# 4.5.1 DESCRIPTION OF STUDY ASSESSMENTS

All patients will be closely monitored for safety and tolerability during all cycles of therapy and at the Study Treatment Discontinuation Visit. Patients should be assessed for toxicity prior to each dose; dosing will occur only if the clinical assessment and local laboratory test values are acceptable. Trastuzumab emtansine will be administered either in q3w cycles (patients with mBC) or qw cycles (patients with mGC) if no additional time is required for resolution of toxicity. Dose delays and dose reductions will be allowed for trastuzumab emtansine as outlined in Section 5.1.5.

If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend that precludes the procedure within the allotted window, the procedure should be performed on the nearest following date (i.e., within 3 business days).

# 4.5.1.1 Medical History and Demographic Data

Medical history includes clinically significant diseases, surgeries, cancer history (including prior cancer therapies and procedures), smoking history, use of alcohol and drugs of abuse, and all medications (e.g., prescription drugs, overthe-counter drugs, herbal/homeopathic remedies, nutritional supplements) used by the patient within 14 days prior to the screening visit.

Demographic data will include age, sex, and self-reported race/ethnicity (unless not allowed per local regulations).

# 4.5.1.2 Vital Signs

Vital signs will include measurements of weight, respiratory rate, heart rate, blood pressure, and temperature. Abnormal or significant changes to vital signs from baseline should be recorded as AEs, if appropriate.

# 4.5.1.3 Physical Examinations

A complete physical examination should include the evaluation of head, eye, ear, nose, and throat; cardiovascular; dermatological; musculoskeletal; respiratory; gastrointestinal; and neurological systems. Changes from baseline abnormalities should be recorded at each subsequent physical examination. New or worsened abnormalities should be recorded as AEs if appropriate.

As part of the tumor assessment, physical examinations should also include the evaluation of the presence and degree of enlarged lymph nodes, hepatomegaly, and splenomegaly.

Limited physical examinations will be symptom-directed.

# 4.5.1.4 Tumor and Response Evaluations

Measurable and unmeasurable disease must be documented at screening and re-assessed at each subsequent tumor evaluation. Tumor assessments with computed tomography (CT) or magnetic resonance imaging (MRI) scans of the chest, abdomen, and pelvis are to be performed as described in Appendix 1, Schedule of Assessment. CT or MRI of the brain and baseline radioisotope bone scan must be obtained at screening. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to first treatment the bone scan does not need to be repeated and non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Tumor assessments should include an evaluation of all known and/or suspected sites of disease, whenever possible. Patients should have lesions selected that can be evaluated at every tumor assessment. The same radiographic procedure used at screening must be used throughout the study (e.g., the same contrast protocol for CT scans). Response assessments will be assessed by the investigator, based on physical examinations, CT or MRI scans, and bone scans using RECIST v. 1.1 (see Appendix 3). In the event a positron emission tomography (PET)/CT scanner is used for tumor assessments, the CT portion of the PET/CT must meet criteria for diagnostic quality. For patients who continue study treatment after isolated brain progression, the frequency of follow-up scans is at the discretion of the investigator.

At the investigator's discretion, CT scans, MRI scans, and/or bone scans may be obtained at any time when clinically indicated or if PD is suspected. If a bone scan cannot be performed during the course of the study because of the unavailability of the Tc-99m isotope, the investigator may choose an alternative imaging modality (see <a href="Appendix 4">Appendix 4</a>).

Radiographic imaging should always be performed rather than clinical examination unless the lesion(s) being followed cannot be imaged but is assessable by clinical examination. In applying RECIST, documentation by color photography including a ruler to estimate the size of the lesion is recommended.

# 4.5.1.5 Laboratory Assessments

#### For Patients with mBC:

## **Local Laboratory Assessments:**

- Hematology, biochemistry, coagulation, urinalysis, and pregnancy testing
- Prospective or retrospective HER2 status. Patients will be enrolled based on local results.

# **Central Laboratory Assessments:**

- Retrospective HER2 status. Retrospective central confirmation will not impact the treatment decisions or primary endpoint of Phase I, Cohort 1 and will be used to validate efficacy analyses in Phase I and to define subgroups for efficacy analyses in the Randomized Phase II part of the study
- PK assays:
- Serum trastuzumab emtansine concentration and total trastuzumab using a validated immunoassay
- Serum capecitabine and 5-FU PK samples
- Plasma concentration of DM1 using a validated liquid chromatography electrospray tandem mass spectrometry (LC-MS/MS) method

#### For Patients with mGC:

#### **Local Laboratory Assessments:**

Hematology, biochemistry, coagulation, urinalysis, and pregnancy testing

### **Central Laboratory Assessments:**

- Prospective HER2 status. Patients will be enrolled based on the central testing results
- PK assays:
- Serum trastuzumab emtansine concentration and total trastuzumab using a validated immunoassay
- Serum capecitabine and 5-FU PK samples
- Plasma concentration of DM1 using a validated LC-MS/MS method

# 4.5.1.6 Electrocardiograms

A 12-lead ECG should be obtained at baseline and be printed and kept with the patient's record.

#### 4.5.1.7 ECOG Performance Status

Performance status will be measured using the ECOG performance status scale (see Appendix 6).

It is recommended, where possible, that a patient's performance status be assessed by the same person throughout the study.

Performance status will be assessed according to the schedule of assessments (see Appendix 1).

### 4.5.1.8 ECHO/MUGA

ECHO is the preferred modality because of the global technetium (Tc-99m) shortage (see Appendix 4). The same method used at screening should be used throughout the study.

# 4.5.2 TIMING OF STUDY ASSESSMENTS

# 4.5.2.1 Screening and Pretreatment Assessments

Written informed consent for participation in the study must be obtained before performing any study-specific screening tests or evaluations. Informed Consent Forms for enrolled patients and for patients who are not subsequently enrolled will be maintained at the study site.

Once the patient has signed the Informed Consent Form, the investigator (or his or her designee) will call the IxRS to obtain the screening number for the patient prior to Cycle 1, Day 1.

Results of standard of care tests or examinations performed prior to obtaining informed consent and within 28 days prior to study start may be used; such tests do not need to be repeated for screening. Patients must have stable LFTs before the first dose of study drug.

All screening evaluations must be completed and reviewed to confirm that patients meet all eligibility criteria before study start. The investigator will maintain a screening log to record details of all patients screened and to confirm eligibility or record reasons for screening failure, as applicable.

Patients in Cohort 1 will not contribute to Phase II; however, they will be followed up until EOS. In the Randomized Phase II part, patients will be randomized in a 1:1 ratio to receive trastuzumab emtansine alone or the combination of trastuzumab emtansine and capecitabine prior to receiving the first dose of study medication.

The IxRS will be available 24 hours a day, 7 days a week. Detailed instructions regarding the IxRS will be provided to each study center. The screening numbers are to be allocated according to the specification document agreed with the IxRS provider.

Please see Appendix 1 for the schedule of screening assessments.

# 4.5.2.2 Assessments during Treatment

#### For Patients with mBC

Scheduled study visits are based on a q3w cycle, with Cycle 1 beginning at Day 1. All visits must occur within ± 3 business days from the scheduled date, unless otherwise noted in the schedule of assessments. All assessments will be performed on the day of the specified visit unless a time window is specified. Assessments scheduled on the day of study treatment administration should be performed prior to study treatment administration unless otherwise noted. If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend, it should be performed on the nearest following date (i.e., within 3 business days).

Local laboratory assessments scheduled for Day 1 of all cycles must be performed within 72 hours prior to study treatment administration unless otherwise specified. Results of local laboratory assessments must be reviewed and the review documented prior to study treatment administration.

Please see Appendix 1 for the schedule of treatment period assessments.

#### For Patients with mGC

Scheduled study visits are based on a qw cycle, with Cycle 1 beginning at Day 1. All visits must occur within  $\pm$  3 business days from the scheduled date, unless otherwise noted in the schedule of assessments. All assessments will be performed on the day of the specified visit unless a time window is specified. Assessments scheduled on the day of study treatment administration should be performed prior to study treatment administration unless otherwise noted. If the timing of a protocol-mandated procedure coincides with a holiday and/or weekend, it should be performed on the nearest following date (i.e., within 3 business days).

Local laboratory assessments scheduled for Day 1 of all cycles must be performed within 72 hours prior to study treatment administration unless otherwise specified. Results of local laboratory assessments must be reviewed and the review documented prior to study treatment administration.

Please see Appendix 1 for the schedule of treatment period assessments.

# 4.5.2.3 Assessments at Study Completion/Early Termination Visit

Patients may remain on study treatment until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor. Patients who discontinue study treatment will be followed up until EOS and will be asked to return to the clinic approximately 28–42 days after the last study treatment administration for the safety follow-up visit.

Please see Appendix 1 for assessments to be performed at the safety follow-up visit.

# 4.5.2.4 Follow-up Assessments

After the Study Treatment Discontinuation Visit, all patients (regardless of reason for discontinuation) will have survival status and anti-cancer therapies recorded and will be followed for all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or dies, or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration.

Patients who discontinue study drugs for any reason other than PD or withdrawal of consent (e.g., an AE) will continue to be followed according to the tumor assessment schedule until withdrawal of consent, death, or EOS, whichever occurs first.

After the study treatment completion/early termination visit, AEs should be followed as outlined in Section 5.5 and 5.6.

Please see Appendix 1 for the schedule of follow-up assessments.

# 4.5.2.5 Assessments at Unplanned Visits

In case unplanned visits are required, electronic Case Report Form (eCRF) pages will be available to report the information collected during those visits.

# 4.6 PATIENT AND STUDY DISCONTINUATION

#### 4.6.1 PATIENT DISCONTINUATION

Patients have the right to withdraw from the study at any time for any reason. The investigator has the right to discontinue a patient from study treatment or from the study for any medical condition that the investigator determines may jeopardize the patient's safety if he or she continues in the study, for reasons of non-compliance (e.g., missed doses, visits), if the patient becomes pregnant, or if the investigator determines it is in the best interest of the patient.

Patients must be withdrawn from study treatment if they become pregnant or experience PD defined using RECIST v. 1.1 (<u>Appendix 3</u>). The exception to this is patients who develop isolated progression in the brain as described in <u>Appendix 3</u>.

Details of discontinuation due to toxicity are given in Section 5.1.

Patients who discontinue from study treatment prematurely for any of the above reasons will continue to be followed according to Section 4.5.2.4 "Follow-Up Assessments". The primary reason for discontinuation must be recorded on the appropriate eCRF page.

# 4.6.2 STUDY DISCONTINUATION

Sections 3.1.1 and 3.2 describe the EOS definition and discontinuation of study treatment. Prior to that, the Sponsor has the right to terminate this study at any time. Reasons for terminating the study may include, but are not limited to, the following:

- The incidence or severity of AEs in this or other studies indicates a potential health hazard to patients
- Patient enrollment is unsatisfactory
- Data recording is inaccurate or incomplete.

# 5. ASSESSMENT OF SAFETY

Overall safety will be assessed on an ongoing basis during the conduct of the study.

# 5.1 SAFETY PLAN

The safety plan for patients receiving trastuzumab emtansine is based on the toxicities of trastuzumab emtansine observed in nonclinical studies; the toxicities related to its components (trastuzumab and maytansine, the parent drug of DM1) observed in clinical studies; and the clinical experience with this molecule in completed and ongoing studies. Please refer to the trastuzumab emtansine and capecitabine (Xeloda®) Investigator's Brochures for the most recent information.

All patients will be monitored closely for toxicity. The important safety issues anticipated in this trial, as well as measures intended to avoid or minimize such toxicities, are outlined in the following sections.

# 5.1.1 RISKS ASSOCIATED WITH TRASTUZUMAB EMTANSINE

Full details regarding the clinical safety of trastuzumab emtansine are presented in Sections 5 and 6 of the Investigator's Brochure.

# 5.1.1.1 Cardiotoxicity

Patients treated with trastuzumab emtansine are at increased risk of developing left ventricular dysfunction. LVEF < 40% has been observed in patients treated with trastuzumab emtansine. Patients without significant cardiac history and with an LVEF  $\ge$  50% determined by ECHO or MUGA scan are eligible for study participation. LVEF will be monitored at screening and regularly throughout the study until the assessment at the safety follow-up visit. Patients with symptomatic cardiac dysfunction will be discontinued from study treatment. Asymptomatic LVEF declines will be handled according to the algorithm shown in Figure 6. Treatment with trastuzumab emtansine has not been studied in patients with LVEF < 50%.

# 5.1.1.2 Hematologic Toxicity (Thrombocytopenia)

Thrombocytopenia, or decreased platelet counts, was reported in patients in clinical trials of trastuzumab emtansine. The majority of these patients had Grade 1 or 2 events ( $\geq 50,000/\text{mm}^3$ ), with the nadir occurring by Day 8 and generally improving to Grade 0 or 1 ( $\geq 75,000/\text{mm}^3$ ) by the next scheduled dose. In clinical trials, the incidence and severity of thrombocytopenia were higher in Asian patients. Severe cases of both non-fatal and fatal hemorrhagic events including central nervous system hemorrhage have been reported in clinical trials with trastuzumab emtansine; these events were independent of the patients' ethnicity. In some of the observed cases the patients were also receiving anti-coagulation therapy. The need for platelet transfusions has been reported.

Patients with thrombocytopenia and on anti-coagulant treatment have to be monitored closely during treatment with trastuzumab emtansine. Platelet counts will be monitored prior to each trastuzumab emtansine dose.

Use of erythropoiesis-stimulating agents will be allowed as consistent with prescribing guidelines. Transfusion of red blood cells and/or platelets will be allowed according to and at the discretion of the treating physician.

# 5.1.1.3 Hepatotoxicity

Hepatotoxicity, predominantly in the form of asymptomatic increases in the concentrations of serum transaminases (Grade 1–4 transaminitis), has been observed in patients while on treatment with trastuzumab emtansine in clinical trials. Transaminase elevations were generally transient. A cumulative effect of trastuzumab emtansine on transaminases has been observed; elevated transaminases improved to Grade 1 or normal within 30 days of the last dose of trastuzumab emtansine in the majority of the patients.

Serious hepatobiliary disorders, including nodular regenerative hyperplasia (NRH) of the liver and some resulting in fatal liver failure, have been observed in patients treated with trastuzumab emtansine in clinical trials. Some of the observed cases may have been confounded by comorbidities and/or concomitant medications with known hepatotoxic potential. Liver function should be monitored before initiation of treatment and each trastuzumab emtansine dose.

Trastuzumab emtansine has not been studied in patients with serum transaminases  $> 2.5 \times \text{ULN}$  or total bilirubin  $> 1.5 \times \text{ULN}$  before initiation of treatment. Trastuzumab emtansine treatment in patients with serum transaminases  $> 3 \times \text{ULN}$  and concomitant total bilirubin  $> 2 \times \text{ULN}$  should be permanently discontinued.

Cases of NRH of the liver have been identified from liver biopsies in patients presenting with signs and symptoms of portal hypertension. NRH was also observed in one fatal case of hepatic failure. NRH is a rare liver condition characterized by widespread benign transformation of hepatic parenchyma into small regenerative nodules; NRH may lead to non-cirrhotic portal hypertension. Diagnosis of NRH can only be confirmed by histopathology. NRH should be considered in patients who develop clinical symptoms of portal hypertension and/or a cirrhosis-like pattern seen on CT scan of the liver but with normal transaminases and no other manifestations of cirrhosis or liver failure following long-term treatment with trastuzumab emtansine. Upon diagnosis of NRH, trastuzumab emtansine treatment must be permanently discontinued.

# 5.1.1.4 Pulmonary Toxicity

Cases of interstitial lung disease (ILD), including pneumonitis, some leading to acute respiratory distress syndrome or fatal outcome, have been reported in clinical trials with trastuzumab emtansine. Signs and symptoms include dyspnea, cough, fatigue, and pulmonary infiltrates. These events may or may not occur as sequelae of infusion reactions. Treatment has included administration of steroids and oxygen, and study drug discontinuation. Patients with dyspnea at rest due to complications of advanced malignancy and comorbidities may be at increased risk of pulmonary events.

Treatment with trastuzumab emtansine has to be permanently discontinued in patients who are diagnosed with ILD or pneumonitis.

# 5.1.1.5 Infusion-related Reactions/Hypersensitivity

Infusion-related reactions characterized by one or more of the following symptoms, flushing, chills, pyrexia, dyspnea, hypotension, wheezing, bronchospasm, and tachycardia may occur with the administration of monoclonal antibodies and have been reported with trastuzumab emtansine. In general, these symptoms were not severe. In most patients, these reactions resolved over the course of several hours to a day after the infusion was terminated. Patients should be observed closely for infusion-related reactions, especially during the first infusion.

Patients should be observed closely for hypersensitivity. Serious, allergic/anaphylactic-like reactions have been observed in clinical trials with treatment of trastuzumab emtansine. Administration of trastuzumab emtansine will be performed in a setting with access to emergency facilities and staff who

are trained to monitor and respond to medical emergencies. Patients will be observed closely for infusion-related/hypersensitivity during and after each trastuzumab emtansine infusion for a minimum of 90 minutes after the first infusion and for a minimum of 30 minutes after subsequent infusions in the absence of infusion-related AEs. Pre-medication is allowed according to standard practice guidelines. In the event of a true hypersensitivity reaction (in which severity of reaction increases with subsequent infusions), trastuzumab emtansine treatment must be permanently discontinued. Patients who experience a Grade  $\geq$  3 allergic reaction or acute respiratory distress syndrome will be discontinued from study treatment.

# 5.1.1.6 Neurotoxicity

DM1, an anti-microtubule agent, can potentially cause peripheral neuropathy. Peripheral neuropathy, mainly Grade 1 and predominantly sensory, has been reported in clinical trials of trastuzumab emtansine. Treatment with trastuzumab emtansine should be temporarily discontinued in patients experiencing Grade 3 or 4 peripheral neuropathy until symptoms resolve or improve to  $\leq$  Grade 2. Patients should be examined for signs of peripheral neuropathy prior to each dose of trastuzumab emtansine. Patients who experience Grade  $\geq$  3 neurotoxicity in the form of peripheral neuropathy that does not resolve to Grade  $\leq$  2 within 42 days after last dose received will be discontinued from study treatment.

## 5.1.1.7 Extravasation

In trastuzumab emtansine clinical studies, reactions secondary to extravasation have been observed. These reactions were usually mild and comprised erythema, tenderness, skin irritation, pain, or swelling at the infusion site. Rare reports of more severe events such as cellulitis, pain (tenderness and burning sensation), and skin irritation have been received as part of the continuing surveillance of trastuzumab emtansine safety. These reactions have been observed more frequently within 24 hours of infusion. Specific treatment for trastuzumab emtansine extravasation is unknown at this time. The infusion site should be closely monitored for possible subcutaneous infiltration during drug administration.

#### 5.1.1.8 Trastuzumab Emtansine Dose Modification

Trastuzumab emtansine dose modifications are described in Section 5.1.5.1.

# 5.1.2 RISKS ASSOCIATED WITH CAPECITABINE

Patients treated with capecitabine should be carefully monitored for toxicity. Most AEs are reversible and do not require permanent discontinuation of therapy (please refer to the Xeloda<sup>®</sup> SmPC for more information).

The spectrum of cardiotoxicity observed with capecitabine is similar to that of other fluorinated pyrimidines. This includes myocardial infarction, angina,
dysrhythmias, cardiac arrest, cardiac failure and electrocardiographic changes. These AEs may be more common in patients with a prior history of coronary artery disease.

Rarely, unexpected, severe toxicity (e.g. stomatitis, diarrhea, mucosal inflammation, neutropenia, and neurotoxicity) associated with 5-FU has been attributed to deficiency of dihydropyrimidine dehydrogenase (DPD) activity. Patients with low or absent DPD activity, an enzyme involved in fluorouracil degradation, are at increased risk for severe, life-threatening, or fatal adverse reactions caused by fluorouracil.

Although DPD deficiency cannot be precisely defined, it is known that patients with certain homozygous or certain compound heterozygous mutations in the *DPYD* gene locus, which can cause complete or near complete absence of DPD enzymatic activity (as determined by laboratory assays), have the highest risk of life-threatening or fatal toxicity<sup>47</sup> and should not be treated with capecitabine. No dose has been proven safe for patients with complete absence of DPD activity.

For patients with partial DPD deficiency (such as those with heterozygous mutations in the *DPYD* gene) and where the benefits of capecitabine are considered to outweigh the risks (taking into account the suitability of an alternative non-fluoropyrimidine chemotherapeutic regimen), these patients must be treated with extreme caution and frequent subsequent monitoring and dose adjustment according to toxicity. There is insufficient data to recommend a specific dose in patients with partial DPD activity as measured by specific test.

In patients with unrecognized DPD deficiency treated with capecitabine, life-threatening toxicities manifesting as acute overdose may occur. In the event of Grade 2–4 acute toxicity, treatment must be discontinued immediately. Permanent discontinuation should be considered based on clinical assessment of the onset, duration, and severity of the observed toxicities.

Capecitabine can induce hand-foot syndrome (palmar-plantar erythrodysesthesia or chemotherapy-induced acral erythema), which is a cutaneous toxicity. Persistent or severe hand-foot syndrome (Grade 2 and above) can eventually lead to loss of fingerprints, which could impact patient identification. For patients receiving capecitabine monotherapy in the metastatic setting, the median time to onset was 79 days (range 11–360 days), with a severity range of Grades 1 to 3. Grade 1 hand-foot syndrome is defined by numbness, dysesthesia/paresthesia, tingling or erythema of the hands and/or feet and/or discomfort which does not disrupt normal activities. Grade 2 is defined as painful erythema and swelling of the hands and/or feet and/or discomfort affecting the patient's activities of daily living (ADL). Grade 3 is defined as moist desquamation, ulceration, blistering or severe pain of the hands and/or feet and/or severe discomfort that causes the patient to be unable to work or perform ADL. If Grade 2 or 3 hand-foot syndrome occurs, administration of capecitabine should be interrupted until the event resolves or decreases in intensity to Grade 1.

Following Grade 3 hand-foot syndrome, subsequent doses of capecitabine should be decreased.

Patients should be carefully monitored for ophthalmological complications such as keratitis and corneal disorders, especially if they have a prior history of eye disorders. Treatment of eye disorders should be initiated as clinically appropriate.

Capecitabine can induce hyperbilirubinemia. Administration of capecitabine should be interrupted if treatment-related elevations in bilirubin of  $> 3.0 \times ULN$  or treatment-related elevations in hepatic aminotransferases (ALT/AST) of Grade  $\geq 2$  occur.

Dehydration may cause acute renal failure, especially in patients with preexisting compromised renal function or when capecitabine is given concomitantly with known nephrotoxic agents. Acute renal failure secondary to dehydration might be potentially fatal.

Capecitabine can induce severe skin reactions such as Stevens-Johnson syndrome and toxic epidermal necrolysis. Capecitabine should be permanently discontinued in patients who experience a severe skin reaction possibly attributable to capecitabine treatment.

Leucovorin affects the pharmacodynamics of capecitabine and may increase the toxicity of capecitabine. This may be relevant in patients receiving folic acid supplementation for folate deficiency due to the similarity between folinic acid and folic acid.

# 5.1.3 RISKS ASSOCIATED WITH TRASTUZUMAB EMTANSINE AND CAPECITABINE COMBINATION

The two DLTs observed in Phase I, Cohort 1 (in mBC) were grade 3 vomiting in one patient and grade 3 elevated AST and ALT in one patient (see Section 3.1.1.2). Both patients were treated at dose level 1 (capecitabine 750 mg/m² bid, days 1–14) in combination with trastuzumab emtansine 3.6 mg/kg q3w). During Phase I in LA/mGC, DLTs for the combination of trastuzumab emtansine and capecitabine will be observed during Cycle 1 (Days 1–21) of this study. The combination treatment must be considered as a new treatment during Cycle 1, and no individual dose reduction will be allowed during Cycle 1; the general DLT rules will be used instead. Interruptions can be made due to toxicities considered by the investigator to be related to capecitabine. Grade 2–4 toxicities should be interrupted until resolved to Grade 0–1. For Grade 4 toxicities, consideration to discontinue treatment with capecitabine will be made with the adjudication of the SC.

#### 5.1.4 DEFINITION OF DOSE-LIMITING TOXICITY

DLTs will be observed during Cycle 1 (Day 1–21). Please refer to the Xeloda® SmPC for recommendations on dose reduction in subsequent cycles.

#### **Definition of DLT:**

#### **Hematologic**

- 1. Uncomplicated Grade 4 thrombocytopenia that does not recover to ≥ 75,000/MI before Day 21
- Thrombocytopenia (any grade) complicated with clinically significant bleeding requiring medical intervention, such as platelet transfusion or cauterization. However, patients with Grade 1 or 2 epistaxis may have cauterization and this should not be considered as a DLT.
- 3. Grade 4 neutropenia lasting > 7 consecutive days
- 4. Febrile neutropenia with an ANC of < 1,000 cells/mm<sup>3</sup>

#### Non-hematologic

- 5. Grade ≥ 3 diarrhea that does not decrease to Grade ≤ 2 after 24 hours of starting recommended anti-diarrheal treatment
- 6. Grade 3 hand-foot syndrome (Grade 4 not applicable)
- 7. Any other treatment-related toxicity Grade ≥ 3 prohibiting the start of the second cycle on Day 22 (3 weeks cycle length plus 1 day)

NOTE: If a Grade 2 event requires a dose delay, it will not be considered as a DLT. However, if the toxicity does not resolve to Grade 1 or baseline by Day 42, this requires discontinuation and will be considered as a DLT.

8. Grade 2 toxicity requiring interruption of treatment for > 14 days

NOTE: Patients experiencing acute early-onset (within 1 week) or unusually severe toxicity of diarrhea, stomatitis, mucosal inflammation, neurotoxicity, neutropenia, or febrile neutropenia with ANC < 500 cells/mm³ during Cycle 1 must be tested for DPD deficiency (a central laboratory will be appointed). The SC will adjudicate in cases of DLTs that are not covered by the existing DLT criteria.

- 9. Having taken < 14 full doses of capecitabine due to toxicity
- 10. Patient not able to receive 100% of the dose level going into Cycle 2, Day 1

#### 5.1.5 MANAGEMENT OF SPECIFIC ADVERSE EVENTS

#### 5.1.5.1 Trastuzumab Emtansine Dose Modification

Patients should be assessed for toxicity prior to each dose; dosing will occur only if the clinical assessment and laboratory test values are acceptable.

Dose delays and reductions are designed to maximize treatment for those who derive clinical benefit from treatment while ensuring patient safety. Dose delays for trastuzumab emtansine-related toxicity other than those specified below (i.e., infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, cardiotoxicity, and ILD or pneumonitis) are as follows:

- If significant trastuzumab emtansine-related toxicities (other than infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, and cardiotoxicity) have not recovered to Grade 1 or baseline, the next scheduled dose may be delayed for up to 42 days from the last dose received. "Significant" and "related" will be based on the judgment of the investigator (in consultation with the Sponsor's Medical Monitor or designee when appropriate). For example, alopecia even if considered related would most likely not be considered to be significant. Fatigue may or may not be considered either related or significant.
- In general, when the significant and related toxicity (or any other toxicity that the investigator chooses to delay dosing for) resolves to Grade 1 or baseline, the patient may resume trastuzumab emtansine if the delay has not exceeded 42 days from the last received dose. Patients should be reevaluated qw during the delay, whenever possible. If dosing resumes, the patient may receive trastuzumab emtansine either at the same dose level as before or at one dose level lower (see Table 2 and Table 3), at the discretion of the investigator. Subsequent cycles should remain the same (q3w or qw), and patients should be assessed for toxicity.
- If a patient requires a dose reduction, dosing will be reduced by one dose level, per Table 2or Table 3. No dose re-escalation will be allowed.
- If toxicity does not resolve within 42 days from the last dose received, the
  patient will be discontinued from study treatment and will be followed for PD
  and survival outcome as described in Section 5.5.
- Patients who experience a Grade 3 or 4 hematologic event should be checked at least weekly for recovery. If values do not recover to baseline or Grade ≤ 1 within 42 days from the last dose received, the patient will be discontinued from study treatment.

Table 2 Dose Reduction for Trastuzumab Emtansine (Patients with mBC)

| Dose Level | q3w Schedule |
|---------------------------------------|---------------------|
| 0 | 3.6 mg/kg |
| - 1 | 3.0 mg/kg |
| - 2 | 2.4 mg/kg |
| Indication for further dose reduction | Off study treatment |

q3w = every 3 weeks

Table 3 Dose Reductions for Trastuzumab Emtansine (Patients with mGC)

| | qw Schedule |
|---------------------------------------|-------------|
| Dose Level | |
| 0 | 2.4 mg/kg |
| - 1 | 2.0 mg/kg |
| - 2 | Off study |
| Indication for further dose reduction | Off study |

qw = weekly

In case of toxicities requiring the discontinuation of trastuzumab emtansine, the patient will be followed-up until the EOS.

Protocol requirements for specific toxicities are outlined below.

### 5.1.5.1.1 Trastuzumab Emtansine Dose Modification for Thrombocytopenia

Platelet counts should be obtained no less frequently than weekly to evaluate recovery whenever any of the events listed below occurs. If platelet counts do not recover to Grade ≤ 1 within 42 days from the last dose received, the patient will be discontinued from study treatment.

No re-escalation of the trastuzumab emtansine dose is allowed.

Note: although complete blood counts with platelets are required within 72 hours prior to study treatment administration at each cycle, the investigator may monitor platelet counts (or any other laboratory test) more frequently as clinically indicated.

In the event of decreased platelet count to Grade 3 ( $< 50,000/mm^3$ ), do not administer trastuzumab emtansine until platelet counts recover to Grade 1 ( $\ge 75,000/mm^3$ ), then treat at the same dose level.

Patients receiving trastuzumab emtansine who experience a first Grade 4 thrombocytopenia event may, after adequate recovery to a platelet count of Grade ≤ 1 or baseline, continue treatment with trastuzumab emtansine at a dose of 3 mg/kg in subsequent treatment cycles. Patients at the 3 mg/kg dose level who experience a Grade 4 thrombocytopenia event may, after adequate recovery as defined above, continue treatment with trastuzumab emtansine at a dose of 2.4 mg/kg in subsequent treatment cycles. Patients who experience a Grade 4 thrombocytopenia event at the 2.4 mg/kg dose level will be discontinued from study treatment. A dose delay of up to 42 days from the patient's last dose received is permitted.

#### 5.1.5.1.2 Trastuzumab Emtansine Dose Modification for Hepatotoxicity

# 5.1.5.1.2.1 Concurrent elevations of ALT/AST and bilirubin meeting Hy's Law laboratory criteria

Regardless of dose level, trastuzumab emtansine must be <u>permanently discontinued</u> in patients with ALT and/or AST > 3 × ULN and concurrent increase of total bilirubin to > 2 × ULN. All relevant hepatic laboratory tests performed (including AST, ALT, total bilirubin, alkaline phosphatase, activated partial thromboplastin time [aPTT], INR, and albumin) will be entered into the clinical database.

#### 5.1.5.1.2.2 Nodular regenerative hyperplasia

Trastuzumab emtansine must be permanently discontinued in patients who are diagnosed with NRH.

# 5.1.5.1.2.3 Transaminase elevations or bilirubin elevation requiring dose adjustment

Patients who experience a Grade 3 elevation of liver function should be checked twice weekly for the recovery of transaminases and/or total bilirubin. If a patient's transaminases and/or total bilirubin do not recover according to Table 4 and Table 5, within 42 days from the patient's last dose received, the patient will be discontinued from study treatment.

No re-escalation of the trastuzumab emtansine dose is allowed.

Table 4 and Table 5 describe the dose modification guidelines for increases in serum bilirubin and transaminases, respectively.

Table 4 Trastuzumab Emtansine Dose Modification: Total Serum Bilirubin

| Grade 2 | Grade 3 | Grade 4 |
|---|---|---|
| (> .5 to ≤ 3 × ULN) | (> 3 to ≤ 10 × ULN) | (> 10 × ULN) |
| Do not administer trastuzumab emtansine until total bilirubin recovers to Grade ≤ 1, and then treat at the same dose level | Do not administer trastuzumab emtansine until total bilirubin recovers to Grade ≤ and then reduce one dose level | Discontinue<br>trastuzumab<br>emtansine |

ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

emtansine

| Grade 2 | Grade 3 | Grade 4 |
|------------------------|-------------------------------|--------------|
| (> 3 to ≤ 5 × ULN) | (> 5 to ≤ 20 × ULN) | (> 20 × ULN) |
| Treat at the same dose | Do not administer trastuzumab | Discontinue |
| level | emtansine until AST/ALT | trastuzumab |

recovers to Grade ≤ 2, and then

Table 5 Trastuzumab Emtansine Dose Modification: Serum ALT or AST

ALT = alanine transaminase; AST = aspartate transaminase; ULN = upper limit of normal. Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

reduce one dose level

#### 5.1.5.1.3 Trastuzumab Emtansine Dose Modification for Neurotoxicity

Patients receiving trastuzumab emtansine who experience Grade 3 or 4 peripheral neuropathy that does not resolve to Grade ≤ 2 within 42 days after the last dose received will be discontinued from study treatment.

#### 5.1.5.1.4 **Trastuzumab Emtansine Dose Modification for Cardiotoxicity**

Patients without significant cardiac history and with a baseline LVEF ≥ 50% as determined by ECHO or MUGA scan are eligible for study participation. Ejection fractions will be monitored during the last week of Cycle 1, Cycle 3 and every third cycle thereafter until the assessment at the safety follow-up visit.

Figure 6 summarizes the management of trastuzumab emtansine on the basis of measured LVEF and changes in LVEF from baseline in patients. If the LVEF is reported as a range, the median of the range should be taken. If an investigator is concerned that an AE may be related to cardiac dysfunction, an additional LVEF measurement may be performed. Trastuzumab emtansine will be discontinued in any patient who develops symptomatic CHF. CHF should be treated and monitored according to standard medical practice.

The decision to stop or continue trastuzumab emtansine should be based on the algorithm shown in Figure 6. Trastuzumab emtansine must be discontinued in all patients for whom a confirmed drop of LVEF to below 40% is documented (with a repeat assessment within 21 days). For patients whose LVEF drops to values between 40% and 45% with an absolute decrease in LVEF of ≥ 10% points from baseline, trastuzumab emtansine should be held. For these patients, the LVEF should be repeated in 21 days, and trastuzumab emtansine should be discontinued if the LVEF has not recovered to within 10% absolute difference below baseline. If clinically significant cardiac dysfunction or cardiac failure develops or persists or if significant medical management is required to maintain ejection fraction, the patient should be discontinued from study treatment.

Figure 6 Algorithm for Continuation and Discontinuation of Trastuzumab Emtansine Based on Left Ventricular Ejection Fraction Assessments in Patients



CHF = congestive heart failure; LVEF = left ventricular ejection fraction.

Note: LVEF assessment results must be reviewed before the next scheduled trastuzumab emtansine infusion.

- <sup>a</sup> LVEF can be repeated within 21 days, and trastuzumab emtansine should be discontinued if LVEF < 40% is confirmed. Trastuzumab emtansine should be held while the repeat LVEF is obtained.
- b After a second consecutive confirmatory result, trastuzumab emtansine should be discontinued if the LVEF is confirmed to be ≥ 10% points below baseline or if medical management was required to correct the LVEF.

# 5.1.5.1.5 Trastuzumab Emtansine Dose Modification/Management for Infusion-related Reactions, Hypersensitivity Reactions

Trastuzumab emtansine treatment should be interrupted in patients with severe infusion-related reactions. Trastuzumab emtansine treatment should be permanently discontinued in the event of life-threatening infusion-related reactions.

Infusion of trastuzumab emtansine should be interrupted for patients who develop dyspnea or clinically significant hypotension.

The infusion should be slowed to  $\leq 50\%$  or interrupted for patients who experience any other infusion-related symptoms. When the patient's symptoms have completely resolved, the infusion may be continued at  $\leq 50\%$  of the rate

prior to the reaction and increased in 50% increments every 30 minutes as tolerated. Infusions may be restarted at the full rate during the next cycle.

Patients who experience trastuzumab emtansine infusion-related temperature elevations to > 38.5°C and/or other infusion-related symptoms may be treated symptomatically with acetaminophen and/or diphenhydramine hydrochloride. Serious infusion-related events manifested by dyspnea, hypotension, wheezing, bronchospasm, tachycardia, reduced oxygen saturation, or respiratory distress should be managed with supportive care, such as oxygen, beta agonists, antihistamines, antipyretics, or corticosteroids at the investigator's discretion. Pre-medication with corticosteroids, antihistamines, and antipyretics may be used before subsequent infusions of trastuzumab emtansine at the investigator's discretion. Patients should be monitored until complete resolution of symptoms. In the event of a true hypersensitivity reaction (i.e., if the severity of reaction increases with subsequent infusions), trastuzumab emtansine treatment must be permanently discontinued. Patients who experience a Grade ≥ 3 hypersensitivity reaction or acute respiratory distress syndrome (ARDS) will be discontinued from the study.

Patients who experience a severe delayed infusion reaction will be discontinued from study treatment.

# 5.1.5.1.6 Trastuzumab Emtansine Dose Modification for Pulmonary Toxicity

Cases of ILD, including pneumonitis (including severe, life-threatening cases) and some leading to ARDS or fatal outcome have been reported with trastuzumab emtansine. Treatment with trastuzumab emtansine has to be permanently discontinued in patients who are diagnosed with ILD or pneumonitis.

#### 5.1.5.1.7 Trastuzumab Emtansine Dose Modification for Extravasation

During the clinical development of trastuzumab emtansine, reactions secondary to extravasation have been observed. These reactions were usually mild and consisted of erythema, tenderness, skin irritation, pain or swelling at the infusion site. Although trastuzumab emtansine is not considered as a vesicant, close monitoring of the infusion site for possible subcutaneous infiltration during drug administration is recommended.

#### 5.1.5.2 Capecitabine Dosage Modification

#### Phase I: Patients with mBC

The dose of capecitabine can be modified from Cycle 2 onwards if considered appropriate by the investigator (please refer to the Xeloda® SmPC for recommendations).

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued in patients with mBC.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

During the Randomized Phase II part of the study, the dose of capecitabine will be modified according to the Xeloda® SmPC.

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued in patients with mBC.

#### Phase I: Patients with mGC

The dose of capecitabine can be modified from cycle 2 onwards if considered appropriate by the investigator (please refer to Xeloda® SmPC for recommendations).

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued (see Section 3.1.1).

#### 5.2 SAFETY PARAMETERS AND DEFINITIONS

Safety assessments will consist of monitoring and recording protocol-defined AEs and SAEs; measurement of protocol-specified hematology, clinical chemistry, and urinalysis variables; measurement of protocol-specified vital signs; and other protocol-specified tests that are deemed critical to the safety evaluation of the study drug(s).

The Sponsor or its designee is responsible for reporting relevant SAEs to the Competent Authority, other applicable regulatory authorities, and participating investigators, in accordance with International Conference on Harmonisation (ICH) guidelines, FDA regulations, European Clinical Trials Directive (Directive 2001/20/EC), and/or local regulatory requirements.

The Sponsor or its designee is responsible for reporting unexpected fatal or life-threatening events associated with the use of the study drug to the regulatory agencies and competent authorities by telephone or fax within 7 calendar days after being notified of the event. The Sponsor or its designee will report other relevant SAEs associated with the use of the study medication to the appropriate competent authorities (according to local guidelines), investigators, and central Institutional Review Boards/Ethics Committees (IRBs/ECs) by a written safety report within 15 calendar days of notification.

#### 5.2.1 ADVERSE EVENTS

According to the ICH Guideline for Good Clinical Practice, an AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any of the following:

 Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product

- Any new disease or exacerbation of an existing disease (a worsening in the character, frequency, or severity of a known condition), except as described in Section 5.3.5.7
- Recurrence of an intermittent medical condition (e.g., headache) not present at baseline
- Any deterioration in a laboratory value or other clinical test (e.g., ECG, X-ray) that is associated with symptoms or leads to a change in study treatment or concomitant treatment or discontinuation from study drug
- AEs that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment (e.g., screening invasive procedures such as biopsies)

# 5.2.2 SERIOUS ADVERSE EVENTS (IMMEDIATELY REPORTABLE TO THE SPONSOR)

A SAE is any AE that meets any of the following criteria:

- Fatal (i.e., the AE actually causes or leads to death)
- Life-threatening (i.e., the AE, in the view of the investigator, places the patient at immediate risk of death)

This does not include any AE that had it occurred in a more severe form or was allowed to continue might have caused death.

- Requires or prolongs inpatient hospitalization (see Section 5.3.5.8)
- Results in persistent or significant disability/incapacity (i.e., the AE results in substantial disruption of the patient's ability to conduct normal life functions)
- Congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug
- Significant medical event in the investigator's judgment (e.g., may jeopardize the patient or may require medical/surgical intervention to prevent one of the outcomes listed above)

The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an AE (rated as mild, moderate, or severe, or according to NCI CTCAE criteria; see Section 5.3.3); the event itself may be of relatively minor medical significance (such as severe headache without any further findings).

Severity and seriousness need to be independently assessed for each AE recorded on the eCRF.

SAEs are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2 for reporting instructions).

### 5.2.3 PROTOCOL-DEFINED EVENTS OF SPECIAL INTEREST/NON-SERIOUS EXPEDITED ADVERSE EVENTS

Non-serious AESIs are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2 for reporting instructions) regardless of the attribution of causality. AESIs for this study include the following:

Potential drug-induced liver injury

Any case of potential drug-induced liver injury as assessed by laboratory criteria for Hy's law will be considered as a protocol-defined event of special interest and will need to be reported to the Sponsor expeditiously.

The following laboratory abnormalities define potential Hy's law cases:

 AST and/or ALT elevations that are > 3 × ULN with concurrent elevation of total bilirubin > 2 × ULN (or clinical jaundice if total bilirubin measures are not available), except in patients with documented Gilbert's syndrome. For patients with Gilbert's syndrome, elevation of direct bilirubin > 2 × ULN should be used instead

Suspected transmission of an infectious agent by the study drug:

 Defined as any organism, virus, or infectious particle (e.g., prion protein transmitting transmissible spongiform encephalopathy), both pathogenic and non-pathogenic. A transmission of an infectious agent may be suspected from clinical symptoms or laboratory findings indicating an infection in a patient exposed to a medicinal product. This term ONLY applies when a contamination of the study drug is suspected, NOT for infections supported by the mode of action, e.g., immunosuppression.

#### 5.2.4 Pregnancy and Contraception

ICH M3 guidance requires precautions to be taken to minimize risk to fetus or embryo when including women of childbearing potential in clinical studies. These precautions include the use of highly effective contraceptive measures, excluding pregnancy at baseline (serum test), continued pregnancy monitoring, and continued pregnancy testing for up to 7 months following last dose of study drug (follow-up period based on PK considerations).

Trastuzumab, a component of trastuzumab emtansine, can cause fetal harm when administered to a pregnant woman; postmarketing case reports indicate that its use during pregnancy increases the risk for oligohydramnios during the second and third trimester. Trastuzumab has also been associated with fetal pulmonary hypoplasia, skeletal abnormalities, and neonatal death (see the Herceptin<sup>®</sup> Package Insert). There are no clinical studies of trastuzumab in pregnant women. Immunoglobulin G (IgG) is known to cross the placental barrier.

Therefore, trastuzumab emtansine should be not used during pregnancy. Women of childbearing potential (who have not undergone surgical sterilization

with a hysterectomy and/or bilateral oophorectomy) and men with partners of childbearing potential must agree to use a highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the patient and/or partner.

Methods of birth control which result in a low failure rate (i.e., < 1% per year) when used consistently and correctly are considered highly effective forms of contraception. The use of the following non-hormonal methods of contraception is acceptable:

- True abstinence, when this is the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, and symptothermal post ovulation methods) and withdrawal are not acceptable methods of contraception.
- Male sterilization (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female patients, the vasectomized male partner should be the sole partner.

Alternatively, use of two of the following effective forms of contraception is acceptable:

- Placement of intrauterine device (IUD) or intrauterine system (IUS).
   Consideration should be given to the type of device being used, as there are higher failure rates for certain types (e.g., steel or copper wire).
- Condom with spermicidal foam/gel/film/cream/suppository
- Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

The use of barrier contraceptives should always be supplemented with the use of a spermicide. The following should be noted:

- Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection.
- However, spermicides alone are ineffective at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

It should be noted that two forms of effective contraception are required. A double barrier method, defined as condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, is acceptable.

Contraception is not a requirement in the case of any of the following:

The female patient or female partner of a male patient is considered not to be
of childbearing potential: if she is postmenopausal, defined by amenorrhea
of ≥ 12 months duration in a woman > 45 years old; or is

- ≥ 40 years of age and has had amenorrhea of ≥ 24 months duration; or has undergone surgical sterilization (hysterectomy and/or bilateral oophorectomy)
- The male patient or male partner of a female patient is surgically sterilized For male patients with a female partner of childbearing potential, cooperation of female partner is required (i.e., use of two forms of contraception as stated above) during the study and for at least 7 months following the last dose of study treatment when a highly effective form of contraception is not appropriate.

Based on PK considerations, contraception must continue for the duration of study treatment and for at least 7 months after the last dose of study treatment.

A female patient or partner of a male patient who becomes pregnant during the study must be instructed to stop taking the study medication and immediately inform the investigator. The investigator should report all pregnancies, including the partners of male patients, to the Sponsor within 24 hours. The investigator should counsel the patient/partner, and discuss the risks of continuing with the pregnancy and the possible effects on the fetus. Monitoring of the patient/partner should continue until conclusion of the pregnancy. Pregnancies occurring up to 7 months after the completion of study medication must also be reported to the investigator. Please refer to Section 5.4.3 for reporting procedures.

It is not known whether trastuzumab or trastuzumab emtansine are excreted in human milk. Maternal IgG is excreted in milk and any of these monoclonal antibodies could harm infant growth and development; therefore, women should be advised to discontinue nursing during trastuzumab emtansine therapy and not to breastfeed for at least 7 months following the last dose of either study drug.

Experimental studies have reported that IgGs are present in both the preejaculate and the seminal plasma.<sup>49</sup> To date, there have been no clinical studies to assess the IgG profile in the pre-ejaculate and seminal plasma in male patients receiving trastuzumab or trastuzumab emtansine. Therefore, as a precaution male patients with female partners of childbearing potential are required to use highly effective form of contraception or use two forms of contraception as outlined above. Similarly, vaginal absorption of trastuzumab emtansine is unknown and therefore male patients with pregnant partners are required to use condoms for the duration of the pregnancy, and then revert to contraceptive methods as outlined above. This is to ensure that the fetus is not exposed to the study medication through vaginal absorption. In addition, sperm or blood donation should not occur for at least 7 months after the last dose of study treatment.

# 5.3 METHODS AND TIMING FOR CAPTURING AND ASSESSING SAFETY PARAMETERS

The investigator is responsible for ensuring that all AEs (see Section 5.2.1 for definition) are recorded on the AE eCRF and reported to the Sponsor in accordance with instructions provided in this section and in Sections 5.4, 5.5, and 5.6.

For each AE recorded on the AE eCRF, the investigator will make an assessment of seriousness (see Section 5.2.2, for seriousness criteria), severity (see Section 5.3.3), and causality (see Section 5.3.4).

#### 5.3.1 ADVERSE EVENT REPORTING PERIOD

Investigators will seek information on AEs at each patient contact. All AEs, whether reported by the patient or noted by study personnel, will be recorded in the patient's medical record and on the AE eCRF.

**After informed consent** has been obtained but **prior to initiation of study drug,** only SAEs caused by a protocol-mandated intervention (e.g., invasive procedures such as biopsies, discontinuation of medications) should be reported (see Section 5.4.2 for instructions for reporting SAEs).

After **initiation of study treatment**, all AEs, regardless of relationship to study drug, will be reported until 28 days after the last administration of study drug. After this period, the investigator is not required to actively monitor for AEs; however, the Sponsor should be notified if the investigator becomes aware of any poststudy SAEs (see Section 5.6).

#### 5.3.2 ELICITING ADVERSE EVENT INFORMATION

A consistent methodology of non-directive questioning should be adopted for eliciting AE information at all patient evaluation time points. Examples of non-directive questions include the following:

"How have you felt since your last clinic visit?"

"Have you had any new or changed health problems since you were last here?"

#### 5.3.3 ASSESSMENT OF SEVERITY OF ADVERSE EVENTS

The AE grading (severity) scale found in the NCI CTCAE (v. 4.0) will be used for assessing AE severity (see Table 6).

Table 6 Adverse Event Severity Grading Scale

| | Severity | Alternate Description <sup>a</sup> |
|---|---|---|
| Grade | | |
| 1 | Mild (apply event-specific NCI CTCAE grading criteria) | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate (apply event-specific NCI CTCAE grading criteria) | Minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental ADL <sup>b</sup> |
| 3 | Severe (apply event-specific NCI CTCAE grading criteria) | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL <sup>c</sup> |
| 4 | Very severe, life-threatening,<br>or disabling (apply event-specific<br>NCI CTCAE grading criteria) | Life-threatening consequences; urgent intervention indicated |
| 5 | Death related to AE | |

ADL = activities of daily living; AE = adverse event; CTCAE = Common Terminology Criteria for Adverse Events; NCI = National Cancer Institute.

The NCI CTCAE v4.0 can be found at:

http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm#ctc\_40

Note: Regardless of severity, some events may also meet regulatory seriousness criteria. Refer to definition of a serious AE (see Section 5.2.2).

- <sup>a</sup> Use these alternative definitions for Grade 1, 2, 3, and 4 events when the observed or reported AE is not in the NCI CTCAE listing.
- b Instrumental ADL refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
- <sup>c</sup> Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

#### 5.3.4 ASSESSMENT OF CAUSALITY OF ADVERSE EVENTS

Investigators should use their knowledge of the patient, the circumstances surrounding the event, temporal relationship of event onset to the initiation of study drug, course of the event considering especially the effects of dose reduction or discontinuation of study drug or reintroduction of study drug (as applicable), known association of the event with the study drug or with similar treatments, known association of the event with the disease under study, presence of risk factors in the patient or use of concomitant medications known to increase the occurrence of the event, presence of non-treatment-related factors that are known to be associated with the occurrence of the event, and an evaluation of any potential alternative causes to determine whether or not an AE is considered to be related to study drugs, indicating "yes" or "no" accordingly. To ensure consistency of causality assessments, investigators should apply the general guidelines outlined in Table 7.

### Table 7 Guidance for Causal Attribution of Adverse Event/Serious Adverse Event

Is the AE/SAE suspected to be caused by the investigational product based on facts, evidence, science-based rationales, and clinical judgment?

YES There is a plausible temporal relationship between the onset of the AE and administration of the investigational product, and the AE cannot be readily explained by the patient's clinical state, intercurrent illness, or concomitant therapies; and/or the AE follows a known pattern of response to the investigational product; and/or the AE abates or resolves upon discontinuation of the investigational product or dose reduction and, if applicable, reappears upon re-challenge.

Investigators should apply facts, evidence, or rationales based on scientific principles and clinical judgment to support a causal/contributory association with an investigational product.

#### NO <u>AEs will be considered related, unless they fulfill the criteria as specified below.</u>

Evidence exists that the AE has an etiology other than the investigational product (e.g., pre-existing medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the AE has no plausible temporal relationship to administration of the investigational product (e.g., cancer diagnosed 2 days after first dose of study drug).

Note: The investigator's assessment of causality for individual AE reports is part of the study documentation process. Regardless of the "Yes" or "No" causality assessment for individual AE reports, the Sponsor will promptly evaluate all reported SAEs against cumulative product experience to identify and expeditiously communicate possible new safety findings to investigators and applicable regulatory authorities. <a href="Attribution of SAEs will be reviewed on an ongoing basis, and may be changed as additional clinical data emerges (e.g., reversibility of AE, new clinical findings in patient with AE, effects of retreatment, AEs in other patients).</a>

In addition to assessing causality with respect to study drugs, investigators should also assess whether other factors (e.g., disease under study, concurrent illness, concomitant medication, or study procedure) may have caused the event, using similar guidance.

The investigator's assessment of causality for individual AE reports is part of the study documentation process. Regardless of the "Yes" or "No" causality assessment for individual AE reports, the Sponsor will promptly evaluate all reported serious AEs against cumulative product experience to identify and expeditiously communicate possible new safety findings to investigators and applicable regulatory authorities.

For patients receiving combination therapy, causality will be assessed individually for each protocol-mandated therapy.

#### 5.3.5 Procedures for Recording Adverse Events

Investigators should use correct medical terminology/concepts when recording AEs on the AE eCRF. Avoid colloquialisms and abbreviations.

There is one eCRF page for recording AEs or SAEs.

Only one AE term should be recorded in the event field on the AE eCRF.

#### 5.3.5.1 Diagnosis *versus* Signs and Symptoms

#### Infusion-related Reactions

AEs that occur during or within 24 hours after study drug infusion should be captured as individual signs and symptoms rather than a diagnosis of allergic reaction or infusion-related reaction. However, a diagnosis has to be captured as an AE if signs and symptoms constitute a diagnosis of allergic reaction/hypersensitivity or infusion-related reaction and are classified as SAEs; all such symptoms have to be described in the narrative (e.g., in the Additional Case Details field of the eCRF).

#### Other Adverse Events

For AEs other than infusion-related reactions, a diagnosis (if known) should be recorded on the AE eCRF rather than individual signs and symptoms (e.g., record only liver failure or hepatitis rather than jaundice, asterixis, and elevated transaminases). However, if a constellation of signs and/or symptoms cannot be medically characterized as a single diagnosis or syndrome at the time of reporting, each individual event should be recorded on the AE eCRF. If a diagnosis is subsequently established, all previously reported AEs based on signs and symptoms should be nullified and replaced by one AE report based on the single diagnosis, with a starting date that corresponds to the starting date of the first symptom of the eventual diagnosis.

#### 5.3.5.2 Adverse Events Occurring Secondary to Other Events

In general, AEs occurring secondary to other events (e.g., cascade events or clinical sequelae) should be identified by their primary cause. For example, if severe diarrhea is known to have resulted in dehydration, it is sufficient to record only diarrhea as an AE or SAE on the eCRF.

However, medically significant AEs occurring secondary to an initiating event that are separated in time should be recorded as independent events on the eCRF. For example, if a severe gastrointestinal hemorrhage leads to renal failure, both events should be recorded separately on the eCRF. All AEs should be recorded separately on the Adverse Event eCRF if it is unclear whether the events are associated.

#### 5.3.5.3 Persistent or Recurrent Adverse Events

A persistent AE is one that extends continuously, without resolution, between patient evaluation time points. Such events should only be recorded once on the AE eCRF. The initial severity of the event should be recorded, and the severity should be updated to reflect the most extreme severity any time the event

worsens. If the event becomes serious, the AE eCRF should be updated to reflect this.

A recurrent AE is one that resolves between patient evaluation time points and subsequently recurs. Each recurrence of an AE should be recorded separately on the AE eCRF.

#### 5.3.5.4 Abnormal Laboratory Values

Only clinically significant laboratory abnormalities that require active management will be recorded as AEs or SAEs on the eCRF (e.g., abnormalities that require study drug dose modification, discontinuation of study treatment, more frequent follow-up assessments, further diagnostic investigation, etc.).

If the clinically significant laboratory abnormality is a sign of a disease or syndrome (e.g., alkaline phosphatase and bilirubin 5 × ULN of normal associated with cholecystitis), only the diagnosis (e.g., cholecystitis) needs to be recorded on the AE eCRF.

If the clinically significant laboratory abnormality is not a sign of a disease or syndrome, the abnormality itself should be recorded as an AE or SAE on the eCRF. If the laboratory abnormality can be characterized by a precise clinical term, the clinical term should be recorded as the AE or SAE. For example, an elevated serum potassium level of 7.0 mEq/L should be recorded as "hyperkalemia."

Observations of the same clinically significant laboratory abnormality from visit to visit should not be repeatedly recorded as AEs or SAEs on the eCRF, unless their severity, seriousness, or etiology changes.

#### 5.3.5.5 Abnormal Vital Sign Values

Not every vital sign abnormality qualifies as an AE. A vital sign result must be reported as an AE if it meets any of the following criteria:

- Is accompanied by clinical symptoms
- Results in a change in study treatment (e.g., dosage modification, treatment interruption, or treatment discontinuation)
- Results in a medical intervention or a change in concomitant therapy
- Is clinically significant in the investigator's judgment

It is the investigator's responsibility to review all vital sign findings. Medical and scientific judgment should be exercised in deciding whether an isolated vital sign abnormality should be classified as an AE.

If a clinically significant vital sign abnormality is a sign of a disease or syndrome (e.g., high blood pressure), only the diagnosis (i.e., hypertension) should be recorded on the Adverse Event eCRF.

Observations of the same clinically significant vital sign abnormality from visit to visit should only be recorded once on the Adverse Event eCRF (see Section 5.3.5.3 for details on recording persistent AEs).

#### 5.3.5.6 Abnormal Liver Function Tests

The finding of an elevated ALT or AST ( $>3 \times$  baseline value) in combination with either an elevated total bilirubin ( $>2 \times$  ULN) or clinical jaundice in the absence of cholestasis or other causes of hyperbilirubinemia is considered to be an indicator of severe liver injury (as defined by Hy's law). Therefore, investigators must report as an AE the occurrence of either of the following:

- Treatment-emergent ALT or AST > 3 × baseline value in combination with total bilirubin > 2 × ULN (of which ≥ 35% is direct bilirubin)
- Treatment-emergent ALT or AST > 3 × baseline value in combination with clinical jaundice

The most appropriate diagnosis or (if a diagnosis cannot be established) the abnormal laboratory values should be recorded on the Adverse Event eCRF (see Section 5.3.5.4) and reported to the Sponsor immediately (i.e., no more than 24 hours after learning of the event), either as an SAE or a non-serious AE of special interest (see Section 5.4.2).

#### 5.3.5.7 Deaths

Deaths that occur during the protocol-specified AE reporting period (see Section 5.3.1), that are attributed by the investigator solely to progression of mBC or mGC should be recorded only on the Study Completion/Early Discontinuation eCRF. All other on-study deaths, regardless of relationship to study drug, must be recorded on the AE eCRF and immediately reported to the Sponsor (see Section 5.4.2). The IDMC will monitor the frequency of death from all causes.

Death should be considered an **outcome** and not a distinct event. The event or condition that caused or contributed to the fatal outcome should be recorded as the single medical concept on the AE eCRF. Generally, only one such event should be reported. If the cause of death is unknown and cannot be ascertained at the time of reporting, "**unexplained death**" should be recorded on the AE eCRF. If the cause of death later becomes available (e.g., after autopsy), "unexplained death" should be replaced by the established cause of death. The term "**sudden death**" should be used only for the occurrence of an abrupt and unexpected death due to presumed cardiac causes in a patient with or without preexisting heart disease, within 1 hour after the onset of acute symptoms or, in the case of an unwitnessed death, within 24 hours after the patient was last seen alive and stable.

During post-study survival follow-up, deaths attributed to progression of mBC or LA/mGC should be recorded only on the Survival eCRF.

#### 5.3.5.8 Pre-Existing Medical Conditions

A pre-existing medical condition is one that is present at the start of this study. Such conditions should be recorded on the Medical and Surgical History eCRF.

A pre-existing medical condition should be recorded as an AE <u>only</u> if the frequency, severity, or character of the condition worsens during the study. When recording such events on the AE eCRF, it is important to convey the concept that the pre-existing condition has changed by including applicable descriptors (e.g., "more frequent headaches" or "worsening gastrointestinal reflux disease").

#### 5.3.5.9 Lack of Efficacy or Clinical Worsening

Events that are clearly consistent with the expected pattern of progression of mBC or LA/mGC should not be recorded as AEs. These data will be captured as efficacy assessment data only. In most cases, the expected pattern of progression will be based on the RECIST criteria. In rare cases, the determination of clinical progression will be based on symptomatic deterioration. However, every effort should be made to document progression using objective criteria. If there is any uncertainty as to whether an event is due to PD, it should be reported as an AE.

#### 5.3.5.10 Hospitalization or Prolonged Hospitalization

Any AE that results in hospitalization or prolonged hospitalization should be documented and reported as a SAE unless specifically instructed otherwise in this protocol.

There are some hospitalization scenarios that do not require reporting as an SAE when there is no occurrence of an AE. These scenarios include a planned hospitalization or prolonged hospitalization to:

- Perform an efficacy measurement for the study
- Undergo a diagnostic or elective surgical procedure for a pre-existing medical condition that has not changed
- Receive scheduled therapy for the target disease of the study

### 5.3.5.11 Adverse Events Associated with an Overdose or Error in Drug Administration

An overdose is the accidental or intentional use of a drug in an amount higher than the dose being studied. An overdose or incorrect administration of study treatment is not itself an AE, but it may result in an AE. All overdose or incorrect administrations of study drug with/without AEs associated should be recorded on the AE eCRF. If the associated AE fulfills seriousness criteria, the event should be reported to the Sponsor immediately (i.e., no more than 24 hours after learning of the event; see Section 5.4.2).

### 5.4 IMMEDIATE REPORTING REQUIREMENTS FROM INVESTIGATOR TO THE SPONSOR

Certain events require immediate reporting to allow the Sponsor to take appropriate measures to address potential new risks in a clinical trial. The investigator must report such events to the Sponsor immediately; under no circumstances should reporting take place more than 24 hours after the investigator learns of the event. The following is a list of events that the investigator must report to the Sponsor within 24 hours after learning of the event, regardless of relationship to study drug:

- SAEs
- Non-serious AESIs
- Pregnancies

The investigator must report new significant follow-up information for these events to the Sponsor immediately (i.e., no more than 24 hours) after becoming aware of the information. New significant information includes the following:

- New signs or symptoms or a change in the diagnosis
- Significant new diagnostic test results
- Change in causality based on new information
- Change in the event's outcome, including recovery
- Additional narrative information on the clinical course of the event

Investigators must also comply with local requirements for reporting SAEs to the local health authority and Institutional Review Board/Ethics Committee (IRB/EC).

#### 5.4.1 EMERGENCY MEDICAL CONTACTS

MEDICAL MONITOR (SPONSOR'S MEDICAL RESPONSIBLE) CONTACT INFORMATION

To ensure the safety of study patients, an Emergency Medical Call Center Help Desk will access the Sponsor Medical Emergency List, escalate emergency medical calls, provide medical translation service (if necessary), connect the investigator with a Sponsor Medical Monitor, and track all calls. The Emergency Medical Call Center Help Desk will be available 24 hours per day, 7 days per week. Toll-free numbers for the Help Desk and Medical Monitor contact information will be distributed to all investigators (see "Protocol Administrative and Contact Information and List of Investigators").

### 5.4.2 REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS AND NON-SERIOUS ADVERSE EVENTS OF SPECIAL INTEREST

For reports of SAEs and non-serious AESIs, investigators should record all case details that can be gathered immediately (i.e., no more than 24 hours) on the AE eCRF and submit the report via the electronic data capture (EDC) system.

A report will be generated and sent to the Sponsor Safety Risk Management by the EDC system.

In the event that the EDC system is unavailable, a paper SAE/Non-Serious AE of Special Interest CRF and Fax Coversheet should be completed and faxed to the Sponsor Safety Risk Management or its designee immediately (i.e., no more than 24 hours) after learning of the event, using the fax numbers provided to investigators (see "Protocol Administrative and Contact Information & List of Investigators"). Once the EDC system is available, all information will need to be entered and submitted via the EDC system.

#### 5.4.3 REPORTING REQUIREMENTS FOR PREGNANCIES

#### **5.4.3.1** Pregnancies in Female Patients

Female patients of childbearing potential will be instructed to immediately inform the investigator if they become pregnant during the study or within 7 months after the last dose of study drug. A Pregnancy Report eCRF should be completed by the investigator immediately (i.e., no more than 24 hours) after learning of the pregnancy and submitted via the EDC system. A Pregnancy Report will automatically be generated and sent to the Sponsor Safety Risk Management. Pregnancy should not be recorded on the AE eCRF. The investigator should have the patient discontinue the study drug and discuss with the patient the risks of the pregnancy and the possible effects on the fetus. Monitoring of the patient should continue until conclusion of the pregnancy.

In the event that the EDC system is unavailable, a Pregnancy Report worksheet and Pregnancy Fax Coversheet should be completed and faxed to the Sponsor Safety Risk Management or its designee immediately (i.e., no more than 24 hours) after learning of the pregnancy, using the fax numbers provided to investigators (see "Protocol Administrative and Contact Information & List of Investigators").

Additional information on any trastuzumab emtansine-exposed pregnancy and infant will be requested by Roche Drug Safety at specific time points (i.e., after having received the initial report, at the end of the second trimester, 2 weeks after the expected date of delivery, and at 3, 6, and 2 months of the infant's life).

Any serious adverse events associated with the pregnancy (e.g., an event in the fetus, an event in the mother during or after the pregnancy, or a congenital anomaly/birth defect in the child) should be reported on the Adverse Event eCRF. In addition, the investigator will submit a Clinical Trial Pregnancy Reporting Form when updated information on the course and outcome of the pregnancy becomes available.

#### 5.4.3.2 Pregnancies in Female Partners of Male Patients

Male patients will be instructed through the Informed Consent Form to immediately inform the investigator if their partner becomes pregnant during the

**Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 4, 23 Mar 2016

102

study or within 7 months after the last dose of study drug. A Pregnancy Report eCRF should be completed by the investigator immediately (i.e., no more than 24 hours) after learning of the pregnancy and submitted via the EDC system. Attempts should be made to collect and report details of the course and outcome of any pregnancy in the partner of a male patient exposed to study drug. The pregnant partner will need to sign an Authorization for Use and Disclosure of Pregnancy Health Information to allow for follow-up on her pregnancy. Once the authorization has been signed, the investigator will update the Pregnancy Report eCRF with additional information on the course and outcome of the pregnancy. An investigator who is contacted by the male patient or his pregnant partner may provide information on the risks of the pregnancy and the possible effects on the fetus, to support an informed decision in cooperation with the treating physician and/or obstetrician.

In the event that the EDC system is unavailable, follow reporting instructions provided in Section 5.4.3.1.

#### 5.4.3.3 Abortions

Any spontaneous abortion should be classified as an SAE (as the Sponsor considers spontaneous abortions to be medically significant events), recorded on the AE eCRF, and reported to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2).

#### 5.4.3.4 Congenital Anomalies/Birth Defects

Any congenital anomaly/birth defect in a child born to a female patient or female partner of a male patient exposed to study drug should be classified as an SAE, recorded on the AE eCRF, and reported to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2).

# 5.5 FOLLOW-UP OF PATIENTS AFTER ADVERSE EVENTS

#### 5.5.1 INVESTIGATOR FOLLOW-UP

The investigator should follow all unresolved AEs and until the events are resolved or stabilized, the patient is lost to follow-up, or it has been determined that the study treatment or participation is not the cause of the AE/SAE. Resolution of AEs and SAEs (with dates) should be documented on the AE eCRF and in the patient's medical record to facilitate source data verification (SDV).

All pregnancies reported during the study should be followed until pregnancy outcome. If the EDC system is not available at the time of pregnancy outcome, follow reporting instructions provided in Section 5.4.3.1.

#### 5.5.2 Sponsor Follow-up

For SAEs, non-serious AESIs, and pregnancies, the Sponsor or a designee may follow-up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details and outcome information (e.g., from hospital discharge summaries, consultant reports, autopsy reports) in order to perform an independent medical assessment of the reported case.

#### 5.6 POST-STUDY ADVERSE EVENTS

At the time of study completion or study discontinuation, the investigator should instruct each patient to report to the investigator any subsequent AEs that the patient's physician believes could be related to prior study drug treatment or study procedures.

The investigator is not required to actively monitor patients for AEs after the end of the AE reporting period (defined as 28 days after the last dose of study drug). However, the Sponsor should be notified if the investigator becomes aware of any death or other SAE occurring after the end of the AE reporting period, regardless of causality.

The investigator should report these events directly to Roche Safety Risk Management via telephone or via facsimile using the Roche Clinical Trial (SAE) Reporting Form.

# 5.7 EXPEDITED REPORTING TO HEALTH AUTHORITIES, INVESTIGATORS, INSTITUTIONAL REVIEW BOARDS, AND ETHICS COMMITTEES

To determine reporting requirements for single AE cases, the Sponsor will assess the expectedness of these events using the following reference documents:

Trastuzumab emtansine and capecitabine Investigator's Brochures

The Sponsor will compare the severity of each event and the cumulative event frequency reported for the study with the severity and frequency reported in the applicable reference document.

Reporting requirements will also be based on the investigator's assessment of causality and seriousness, with allowance for upgrading by the Sponsor as needed.

The IDMC will closely monitor the incidence of these expected events during the study. An aggregate report of any clinically relevant imbalances that do not favor the test product will be submitted to health authorities.

# 6. <u>STATISTICAL CONSIDERATIONS AND ANALYSIS</u> PLAN

The design of this study includes: Phase I, Randomized Phase II and different cohorts. Corresponding analyses as described in the protocol will be performed when all data for a particular cohort and study phase are collected and cleaned.

#### Phase I: Patients with mBC:

Enrollment into Cohort 1, patients with HER2-positive mBC, will open first.

Enrolled patients will receive study drug until Investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

Patients randomized in Phase II will receive study drug until investigatorassessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.

The primary analysis of BOR will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever comes first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after the randomization of the first patient.

The EOS analysis will include an updated analysis of BOR, which will be done in a purely exploratory manner.

#### Phase I: Patients with mGC:

Once the MTD is established for Cohort 1, enrollment of patients with HER2-positive and LA/mGC into Cohort 2 will be opened.

Enrolled patients will receive study drug until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.

#### 6.1 DETERMINATION OF SAMPLE SIZE

#### Sample Size for Phase I: mBC

This part will be based on a classical 3 plus 3 Phase I design. A minimum of 6 and up to 18 patients will be enrolled into Cohort 1. There is no formal sample size estimation for this part.

### Sample Size for Randomized Phase II: Exploration of Efficacy and Safety in mBC

The sample size for the primary endpoint BOR is based on a Fisher's exact test with an alpha level of 5% (one-sided),<sup>50,51</sup> power of 70% and the clinical assumption of a BOR rate of 43% with trastuzumab emtansine alone and 62.5% with the combination of trastuzumab emtansine and capecitabine. Approximately 160 patients (approximately 80 patients in each treatment group), including a 15% withdrawal rate, will be randomized with a 1:1 ratio to trastuzumab emtansine alone or the combination of trastuzumab emtansine and capecitabine.

An expected BOR rate of 43.6% (95% CI: 38.6%–48.6%) for patients receiving trastuzumab emtansine alone was chosen based on previously published data for T-DM1 in patients with unresectable, locally advanced or mBC previously treated with a taxane and trastuzumab (EMILIA study).<sup>27</sup>

The BOR rates for patients treated with the combination of T-DM1 and capecitabine were chosen based on recent results from other combination studies of T-DM1 plus chemotherapy or trastuzumab plus capecitabine. Response rates were based on those observed in patients with HER2-positive mBC in a Phase Ib/IIa study (BP22752) that compared the combination of trastuzumab emtansine with docetaxel, with or without pertuzumab (ORR: 76% [95% CI: 53%–92%]), and also in a Phase II study that compared the combination of trastuzumab with docetaxel, with or without capecitabine (ORRs: 72.7% [95% CI: 63.4%–80.8%] and 70.5% [95% CI: 61.2%–78.8%]).<sup>41</sup>

Increased BOR rates for the combination treatment compared with single-agent trastuzumab emtansine are in line with previously published results of a randomized Phase III study in patients with locally advanced or mBC treated with the combination of trastuzumab with capecitabine *versus* capecitabine alone (ORR: 48.1% *versus* 27.0%, odds ratio = 2.50, p = 0.0115).9

The estimation of sample size was performed by Nquery<sup>®</sup> and EAST<sup>®</sup> programs.

#### **Stratification Factors**

The following stratification factor will be implemented in the Randomized Phase II of the study:

 Number of prior lines of treatment for metastatic disease (≤1 or >1; excluding single-agent hormones)

A treatment line is any regimen given to a patient from treatment initiation until confirmed PD.

#### Sample Size for Phase I: mGC

This part will be based on a classical 3 plus 3 Phase I design. From 3 to 12 patients might be enrolled into Cohort 2. There is no formal sample size estimation for this part.

#### 6.2 SUMMARIES OF CONDUCT OF STUDY

#### Phase I: Patients with mBC

Due to the small sample size, per-protocol (PP) population will not be defined for the Phase I, Cohort 1.

Major protocol violations will be summarized by treatment dosage. Median followup will be estimated for Phase I, Cohort 1.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

For the Randomized Phase II part of the study, a PP population will be defined (Section 6.4).

Patient enrollment, duration of follow-up, discontinuation from study treatment and study, and reasons for study discontinuation will be summarized by treatment group for all randomized patients. In addition, major protocol violations will be summarized by treatment arm.

#### Phase I: Patients with LA/mGC

Due to the small sample size, a PP population will not be defined for the Phase I, Cohort 2.

Major protocol violations will be summarized by treatment dosage. Median followup will be estimated for Phase I, Cohort 2.

### 6.3 SUMMARIES OF TREATMENT GROUP COMPARABILITY

#### Phase I: mBC

As Phase I is the MTD-Finding part of the study, there are no treatment group comparisons for this part of the study.

Demographics, medical history, and baseline characteristics will be summarized. Continuous variables will be summarized using median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range. Categorical variables will be summarized by the number and percentage of patients for each treatment dosage.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

The Randomized Phase II part of the study is designed to explore the efficacy and safety of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine alone.

Demographics, medical history, and baseline characteristics will be summarized. Continuous variables will be summarized using median, mean, standard

### **Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 4, 23 Mar 2016

107

deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range. Categorical variables will be summarized by the number and percentage of patients for each treatment group.

#### Phase I: mGC

As Phase I is the MTD-Finding part of the study, there are no treatment group comparisons for this part of the study.

Demographics, medical history and baseline characteristics will be summarized. Continuous variables will be summarized using median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range. Categorical variables will be summarized by the number and percentage for each treatment dosage.

#### 6.4 EFFICACY ANALYSES

#### Phase I, Cohort 1: mBC

The main analysis population will be the DLT-evaluable population as defined in Section 6.5.

#### Randomized Phase II: Exploration of Efficacy in mBC

The main analysis population for the efficacy analysis will be the intent-to-treat population (ITT), which will include all patients in the Randomized Phase II part of the study. The PP population will include all ITT patients who have at least one post-baseline tumor assessment during the Phase II part and no major protocol violations, which will be defined in the statistical analysis plan (SAP).

#### Phase I, Cohort 2: mGC

The main analysis population will be the DLT-evaluable population as defined in Section 6.5.

#### 6.4.1 PRIMARY EFFICACY ENDPOINT

#### Phase I, Cohort 1: Patients with mBC

The primary objectives are defining the MTD and establishing the safety profile. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination.

ORR, as a main efficacy endpoint, will be assessed via BOR rate. The BOR is defined as the best response recorded from the date of enrollment until PD, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

#### Randomized Phase II: Exploration of Efficacy in mBC

The primary efficacy endpoint for the Randomized Phase II part of the study is the ORR as assessed via BOR. The BOR is defined as the best response recorded from the start or randomization into the Phase II part of the study and until PD, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. To be assigned a status of PR or CR, i.e., to be a responder, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 28 days after the criteria for response are first met, i.e., patients need to have two consecutive assessments of PR or CR.

The primary hypothesis of interest when comparing ORR – as assessed via BOR – between the two treatment groups (combination of trastuzumab emtansine and capecitabine *versus* trastuzumab emtansine alone) is:

- H0: π TDM1 = π trastuzumab emtansine + capecitabine where π trastuzumab emtansine is BOR in TDM and trastuzumab emtansine + capecitabine is BOR in trastuzumab emtansine + capecitabine
- H: trastuzumab emtansine trastuzumab emtansine + capecitabine

The number and proportions of responders and non-responders (based on BOR) together with 90% Clopper-Pearson CIs will be presented for each treatment group.

The difference in BOR between treatment groups will be displayed with associated 90% CIs using the Hauck-Anderson approach and p-values for the Fisher's exact test.

Logistic analysis will be used to assess the influence of the stratification factor and baseline covariates in an exploratory manner.

The primary analysis of BOR will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever comes first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after the randomization of the first patient.

#### Phase I, Cohort 2: Patients with LA/mGC

The primary objectives are defining the MTD and establishing the safety profile. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination.

ORR, as a main efficacy endpoint, will be assessed via BOR rate. The BOR is defined as the best response recorded from the date of enrollment until PD, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

#### 6.4.2 SECONDARY EFFICACY ENDPOINTS

#### Phase I, Cohort 1: mBC

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### Randomized Phase II: Exploration of Efficacy in mBC

The secondary efficacy endpoints for the Randomized Phase II will be:

- TTR
- DoR
- TTP
- TTF
- PFS
- CBR
- OS

TTR is defined as the time from randomization to first documentation of confirmed PR or CR (whichever occurs first). Patients who do not have a confirmed response will be censored at the date of the last tumor assessment.

DoR is defined as the period from the date of first recorded PR or CR until the date of PD or death from any cause. Patients with no documented progression after CR or PR will be censored at the last date at which they are known to have had the CR or PR. The method for handling censoring is the same as described for PFS below. Only patients with a BOR of CR or PR (i.e., responders) will be included in the analysis of DoR.

For patients with a BOR of CR or PR, TTR is defined as the time from randomization to the date of first CR or PR. The censoring rules will be similar to those of the PFS.

TTP is defined as time from randomization to the first occurrence of PD. Patients who have not progressed at the time of study completion (including patients who have died before PD) or who are lost to follow-up are censored at the date of the last tumor assessment.

TTF is defined as time from randomization until treatment failure, i.e., to PD, death, withdrawal due to AE or laboratory abnormality, or refusal of treatment. Patients who do not experience any of the above events while on study will be censored on the day of their last tumor assessment.

PFS is defined as the time from randomization until the first documented progression of disease or death from any cause, whichever occurs first. Patients with no PFS events will be censored at the time of the last evaluable tumor

assessment. Patients with no post-baseline tumor assessment will be censored at the time of randomization plus 1 day.

OS is defined as the time from randomization until the date of death, regardless of the cause of death. Patients who are alive at the time of data cut-off will be censored at the date of the last follow-up assessment.

Estimates for the survivor function of both treatment groups for TTR, DoR, TTP, TTF, and OS will be obtained by using the Kaplan-Meier method. HRs and associated 90% CIs will be estimated from non-stratified and stratified (based on the stratification factor) Cox regression models.

CBR includes patients whose best (confirmed) response was PR, CR or SD that lasted at least 6 months. CBR will be summarized in a similar way to the primary efficacy endpoint, ORR as assessed by BOR.

#### Phase I, Cohort 2: mGC

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### 6.5 SAFETY ANALYSES

#### Safety Population Phase I, Cohort 1: mBC

The DLT-evaluable population is defined as all enrolled and treated patients who have not experienced any major protocol violation (including violation of the inclusion and exclusion criteria) and completed Cycle 1.

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

The safety population (SP) will include all patients who received at least one dose of study medication during Phase I. Safety endpoints will be summarized by treatment dosage.

Safety parameters for this part of the study will be summarized by treatment dose. The summaries of AEs, SAEs, AEs that caused discontinuation from the study treatment and/or study, and AESIs will be analyzed in a similar way to AEs in Phase II.

The incidence of AEs and SAEs will be summarized according to the primary SOC and, within each SOC, by MedDRA preferred term. Based on the safety profile of trastuzumab emtansine, time to onset of the first episode of any AESI described in Section 5 will also be summarized via Kaplan-Meier estimates. Additional summaries by frequency tables will also be provided for the AESIs. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry will be presented in shift tables of NCI-CTC grade at baseline *versus* worst grade during treatment for Phase I, Cohort 2, and overall.

LVEF will be summarized over time using mean, median and range (minimum and maximum) and will be presented graphically.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### Randomized Phase II: Exploration of Safety in mBC

The SP will include all patients who received at least one dose of study medication during the Randomized Phase II part of the study. Safety endpoints will be summarized by treatment group.

Safety endpoints during Phase II will be assessed via total AEs, Grade ≥3 AEs, SAEs, AESIs (as described in Section 5), fatal AEs and their causes, events to monitor, premature withdrawal from study medication and/or study, laboratory parameters, LVEF, exposure to study medication, concomitant medications, ECOG performance status, and physical examination.

The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by the Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Based on the safety profile of trastuzumab emtansine, time to onset of the first episode of any AESI described in Section 5 will also be summarized via Kaplan-Meier estimates. Additional summaries by frequency tables will be provided for the AESIs. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology, and biochemistry will be presented in shift tables of NCI-CTCAE grade at baseline *versus* worst grade during treatment for the Randomized Phase II part of the study.

LVEF will be summarized over time using mean, median and range (minimum and maximum) and will be presented graphically.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations, will be analyzed in a similar way. The exposure to study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### Safety Population Phase I, Cohort 2: LA/mGC

The DLT-evaluable population is defined as all enrolled and treated patients who have not experienced any major protocol violation (including violation of the inclusion and exclusion criteria) and have completed Cycle 1.

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

The SP will include all patients who received at least one dose of study medication during Phase I. Safety endpoints will be summarized by treatment dosage.

Safety parameters will be analyzed in a similar way to safety parameters in Phase I, Cohort 1: mBC.

#### 6.6 PHARMACODYNAMIC ANALYSES

No pharmacodynamic analyses are planned for this study.

#### 6.7 PHARMACOKINETIC ANALYSES

#### For Phase I only (Patients with mBC and LA/mGC):

The following PK parameters of trastuzumab emtansine, capecitabine and their metabolites (including but not limited to those listed below) will be determined only in the Phase I part of the study for Cohort 1 and Cohort 2 in all patients who receive study treatment using either non-compartmental and/or population methods, if data allow:

- Serum concentrations of trastuzumab emtansine (conjugate) and total trastuzumab
- Plasma concentrations of DM1, capecitabine and its active metabolite 5-FU
- Total exposure (e.g., AUC)
- C<sub>max</sub>
- CL
- V<sub>d</sub>
- T<sub>1/2</sub>

The PK of trastuzumab emtansine, total trastuzumab and DM1 will be compared with historical single-agent PK data to evaluate the potential effect of capecitabine on the PK of trastuzumab emtansine and related analytes. The PK of capecitabine and its active metabolite 5-FU in Cycle 1 (in the absence of trastuzumab emtansine) will be compared with the PK of Cycle 2 (in the

presence of trastuzumab emtansine) to evaluate the potential effect of trastuzumab emtansine on the PK of capecitabine and 5-FU.

All PK parameters will be listed and tabulated by treatment dose and by Cohort. Descriptive summary statistics including arithmetic mean, geometric mean (e.g., AUC and  $C_{max}$ ), median, range, s.d., and coefficient of variation will be presented for each cohort. Nonlinear mixed effects modeling will also be used; details will be presented in the SAP.

PK samples can be obtained ad hoc in case of a SAE or unexpected toxicities which may suggest a potential drug-drug interaction.

#### 6.8 EXPLORATORY ANALYSES

For all patients with mBC (Phase I, cohort 1; Phase II Exploration of Efficacy and Safety in mBC), a retrospective central confirmation of the HER2 status will be done. Further exploratory analysis for HER2-positive patients (based on central confirmation) will be done for selected endpoints such as BOR and safety endpoints (AEs, SAEs, Grade ≥ 3 AEs, and AESIs).

### For the Randomized Phase II only: Exploration of Efficacy and Safety in Patients with mBC:

Subgroup analysis for BOR, safety endpoints (AEs, SAEs, Grade  $\geq$  3 AEs, and AESIs) in Phase II will be presented for: elderly *versus* younger patients, patients with ECOG 0–1 *versus* ECOG 2, and patients with  $\leq$  versus > prior treatment regimen for metastatic disease.

More details about subgroups will be provided in the SAP.

#### **Pharmacoeconomic Endpoint:**

The resource expenditure due to hospitalizations that are not study-defined evaluations while on study treatment will be evaluated. The number of hospital visits, number of days admitted, and type of visits (emergency department *versus* inpatient care) will be collected. The reason for admission (PD *versus* AE) will also be assessed.

#### 6.9 INTERIM ANALYSES

There is no formal efficacy interim analysis.

However, an IDMC will recommend whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 25, 75, and 150 patients have received at least 3 cycles (Cycle 3 Day 21) of treatment in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the course of the Randomized Phase II of the study or as requested.

Efficacy data will be provided only if required by the IDMC to estimate the riskbenefit balance for the patients. Further details on the function and logistics of the IDMC will be provided in the IDMC Charter.

#### 7. <u>DATA COLLECTION AND MANAGEMENT</u>

#### 7.1 DATA QUALITY ASSURANCE

The Sponsor will be responsible for data management of this study, including quality checking of the data. Data entered manually will be collected via EDC using eCRFs. The sites will be responsible for data entry into the EDC system. In the event of discrepant data, the Sponsor will request data clarification from the sites, which the sites will resolve electronically in the EDC system.

The Sponsor will produce an EDC Study Specification document that describes the quality checking to be performed on the data. Central laboratory data and other electronic data will be sent directly to the Sponsor, using the Sponsor's standard procedures to handle and process the electronic transfer of these data.

eCRFs and correction documentation will be maintained in the EDC system's audit trail. System backups for data stored by the Sponsor and records retention for the study data will be consistent with the Sponsor's standard procedures.

#### 7.2 ELECTRONIC CASE REPORT FORMS

eCRFs are to be completed using a Sponsor-designated EDC system. Sites will receive training and have access to a manual for appropriate eCRF completion. eCRFs will be submitted electronically to the Sponsor and should be handled in accordance with instructions from the Sponsor.

All eCRFs should be completed by designated, trained site staff. eCRFs should be reviewed and electronically signed and dated by the investigator or a designee.

At the end of the study, the investigator will receive patient data for his or her site in a readable format on a compact disc that must be kept with the study records. Acknowledgment of receipt of the compact disc is required.

#### 7.3 SOURCE DATA DOCUMENTATION

Study monitors will perform ongoing SDV to confirm that critical protocol data (i.e., source data) entered into the eCRFs by authorized site personnel are accurate, complete, and verifiable from source documents.

Source documents (paper or electronic) are those in which patient data are recorded and documented for the first time. They include, but are not limited to, hospital records, clinical and office charts, laboratory notes, memoranda, patient-reported outcomes, evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies of transcriptions that are
certified after verification as being accurate and complete, microfiche, photographic negatives, microfilm or magnetic media, X-rays, patient files, and records kept at pharmacies, laboratories, and medico-technical departments involved in a clinical trial.

Source documents that are required to verify the validity and completeness of data entered into the eCRFs must not be obliterated or destroyed.

To facilitate SDV, the investigators and institutions must provide the Sponsor with direct access to applicable source documents and reports for trial-related monitoring, Sponsor audits, and IRB/EC review. The investigational site must also allow inspection by applicable health authorities.

### 7.4 USE OF COMPUTERIZED SYSTEMS

When clinical observations are entered directly into an investigational site's computerized medical record system (i.e., in lieu of original hardcopy records), the electronic record can serve as the source document if the system has been validated in accordance with health authority requirements pertaining to computerized systems used in clinical research. An acceptable computerized data collection system (for clinical research purposes) would be one that (1) allows data entry only by authorized individuals; (2) prevents the deletion or alteration of previously entered data and provides an audit trail for such data changes (e.g., modification of file); (3) protects the database from tampering; and (4) ensures data preservation.

In collaboration with the study monitor, Sponsor's Quality Assurance group may assist in assessing whether electronic records generated from computerized medical record systems used at investigational sites can serve as source documents for the purposes of this protocol.

If a site's computerized medical record system is not adequately validated for the purposes of clinical research (as opposed to general clinical practice), applicable hardcopy source documents must be maintained to ensure that critical protocol data entered into the eCRFs can be verified.

### 7.5 RETENTION OF RECORDS

U.S. FDA regulations (21 Code of Federal Regulations §312.62[c]) and the ICH Guideline for Good Clinical Practice (GCP) (see Section 4.9 of the guideline) require that records and documents pertaining to the conduct of this study and the distribution of investigational drug, including eCRFs, Consent Forms, laboratory test results, and medication inventory records, must be retained by the Principal Investigator for 2 years after the last marketing application approval in an ICH region or after at least 2 years have elapsed since formal discontinuation of clinical development of the investigational product. All state and local laws for retention of records also apply.

No records should be disposed of without the written approval of the Sponsor. Written notification should be provided to the Sponsor for transfer of any records to another party or moving them to another location.

For studies conducted outside the United States under a U.S. Investigational New Drug (IND) application, the Principal Investigator must comply with the record retention requirements set forth in the U.S. FDA IND regulations and the relevant national and local health authorities, whichever is longer.

### 8. ETHICAL CONSIDERATIONS

### 8.1 COMPLIANCE WITH LAWS AND REGULATIONS

This study will be conducted in full conformance with the ICH E6 guideline for GCP and the principles of the Declaration of Helsinki, or the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual. The study will comply with the requirements of the ICH E2A guideline (Clinical Safety Data Management: Definitions and Standards for Expedited Reporting). Studies conducted in the United States or under a U.S. IND application will comply with U.S. FDA regulations and applicable local, state, and federal laws. Studies conducted in the European Union (EU)/European economic area (EEA) will comply with the EU Clinical Trial Directive (2001/20/EC).

### 8.2 INFORMED CONSENT

Sponsor's Sample Informed Consent Form will be provided to each site. If applicable, it will be provided in a certified translation of the local language. The Sponsor or its designee must review and approve any proposed deviations from the Sample Informed Consent Form or any alternate Consent Forms proposed by the site before IRB/EC submission. The final IRB/EC-approved Consent Forms must be provided to the Sponsor for health authority submission purposes according to local requirements.

The Consent Form must be signed and dated by the patient or the patient's legally authorized representative before his or her participation in the study. The case history or clinical records for each patient shall document the informed consent process and that written informed consent was obtained prior to participation in the study.

A copy of each signed Consent Form must be provided to the patient or the patient's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

All signed and dated Consent Forms must remain in each patient's study file and must be available for verification by study monitors at any time.

The Informed Consent Form should be revised whenever there are changes to procedures outlined in the informed consent or when new information becomes available that may affect the willingness of the patient to participate.

For any updated or revised Consent Forms, the case history for each patient shall document the informed consent process and that written informed consent was obtained for the updated/revised Consent Form for continued participation in the study. The final revised IRB/EC-approved Informed Consent Form must be provided to the Sponsor for regulatory purposes.

If the site uses a separate Authorization Form for patient authorization to use and disclose personal health information under the U.S. Health Insurance Portability and Accountability Act (HIPAA) regulations, the review, approval, and other processes outlined above apply except that IRB/IEC review and approval may not be required per study site policies.

# 8.3 INSTITUTIONAL REVIEW BOARD OR ETHICS COMMITTEE

This protocol, the Informed Consent Forms, any information to be given to the patient, and relevant supporting information must be submitted to the IRB/EC by the Principal Investigator and reviewed and approved by the IRB/EC before the study is initiated. In addition, any patient enrollment materials must be approved by the IRB/EC.

The Principal Investigator is responsible for providing written summaries of the status of the study to the IRB/EC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC. Investigators are also responsible for promptly informing the IRB/EC of any protocol amendments.

In addition to the requirements to report protocol-defined AEs to the Sponsor, investigators are required to promptly report to their respective IRB/EC all unanticipated problems involving risk to human patients. Some IRBs/ECs may want prompt notification of all SAEs, whereas others require notification only about events that are serious, assessed to be related to study treatment, and are unexpected. Investigators may receive written IND safety reports or other safety related communications from the Sponsor. Investigators are responsible for ensuring that such reports are reviewed and processed in accordance with regulatory requirements and with the policies and procedures established by their IRB/EC and archived in the site's study file.

### 8.4 CONFIDENTIALITY

The Sponsor maintains confidentiality standards by coding each patient enrolled in the study through assignment of a unique patient identification number. This means that patient names are not included in data sets that are transmitted to any Sponsor location.

Patient medical information obtained by this study is confidential and may only be disclosed to third parties as permitted by the Informed Consent Form (or separate authorization for use and disclosure of personal health information) signed by the patient, unless permitted or required by law.

Medical information may be given to a patient's personal physician or other appropriate medical personnel responsible for the patient's welfare, for treatment purposes.

Data generated by this study must be available for inspection upon request by representatives of the U.S. FDA and other national and local health authorities, the Sponsor monitors, representatives, and collaborators, and the IRB/EC for each study site, as appropriate.

### 8.5 FINANCIAL DISCLOSURE

Investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate health authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

# 9. <u>STUDY DOCUMENTATION, MONITORING, AND ADMINISTRATION</u>

### 9.1 STUDY DOCUMENTATION

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented, including but not limited to the protocol, protocol amendments, Informed Consent Forms, and documentation of IRB/EC and governmental approval. In addition, at the end of the study, the investigator will receive the patient data, which includes an audit trail containing a complete record of all changes to data.

### 9.2 SITE INSPECTIONS

Site visits will be conducted by the Sponsor or an authorized representative for inspection of study data, patients' medical records, and eCRFs. The investigator will permit national and local health authorities, the Sponsor monitors, representatives, and collaborators, and the IRBs/ECs to inspect facilities and records relevant to this study.

### 9.3 ADMINISTRATIVE STRUCTURE

The study will have a SC, IDMC, central laboratory, IxRS, eCRF, and will be conducted by a contract research organization (CRO) together with the Sponsor.

## 9.4 PUBLICATION OF DATA AND PROTECTION OF TRADE SECRETS

The results of this study may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the Sponsor prior to submission. This allows the Sponsor to protect proprietary information and to provide comments based on information from other studies that may not yet be available to the investigator.

The Sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter trials only in their entirety and not as individual center data. In this case, a coordinating investigator will be designated by mutual agreement.

Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements. Any formal publication of the study in which contribution the Sponsor personnel exceeded that of conventional monitoring will be considered as a joint publication by the investigator and the appropriate the Sponsor personnel.

Any inventions and resulting patents, improvements, and/or know-how originating from the use of data from this study will become and remain the exclusive and unburdened property of the Sponsor, except where agreed otherwise.

### 9.5 PROTOCOL AMENDMENTS

Any protocol amendments will be prepared by the Sponsor. Protocol amendments will be submitted to the IRB/EC and to regulatory authorities in accordance with local regulatory requirements.

Approval must be obtained from the IRB/EC and regulatory authorities (as locally required) before implementation of any changes, except for changes necessary to eliminate an immediate hazard to patients or changes that involve logistical or administrative aspects only (e.g., change in Medical Monitor or contact information).

### 10. REFERENCES

- International Agency for Research on Cancer. World Health Organization. GLOBOCAN 2012: Estimated cancer incidence, mortality and prevalence worldwide in 2012. http://globocan.iarc.fr/Pages/fact\_sheets\_cancer.aspx (accessed 16 May 2014).
- 2. Sundaresan S, Penuel E, Sliwkowski MX. The biology of human epidermal growth factor receptor 2. Curr Oncol Rep 1999; 1:16–22.
- 3. Slamon DJ, Clark GM, Wong SG, et al. Human breast cancer; correlation of relapse and survival with amplification of the HER2/neo oncogene. Science 1987; 235:177–82.
- Slamon DJ, Leyland-Jones B, Shak S, et al. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med 2001; 344:783–92.
- 5. Marty M, Cognetti F, Maraninchi D, et al. Randomized Phase II trial of the efficacy and safety of trastuzumab combined with docetaxel in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer administered as first-line treatment: the M77001 study group. J Clin Oncol 2005; 23:4265–74.
- 6. Spector NL, Xia W, Burris H 3<sup>rd</sup>, et al. Study of the biologic effects of lapatinib, a reversible inhibitor of ErbB1 and ErbB2 tyrosine kinases, on tumor growth and survival pathways in patients with advanced malignancies. J Clin Oncol 2005; 23:2502–12.
- 7. Austin CD, De Mazière AM, Pisacane PI, et al. Endocytosis and sorting of ErbB2 and the site of action of cancer therapeutics trastuzumab and geldanamycin. Mol Biol Cell 2004; 15:5268–82.
- 8. Baselga J, Cortés J, et al; CLEOPATRA Study Group. Pertuzumab plus trastuzumab plus docetaxel for metastatic breast cancer. N Engl J Med 2012;366(2):109-19.
- 9. von Minckwitz G, du Bois A, Schmidt M, et al. Trastuzumab beyond progression in human epidermal growth factor receptor 2-positive advanced breast cancer: a german breast group 26/breast international group 03-05 study. J Clin Oncol 2009;27(12):1999-2006.
- 10. Geyer CE, Forster J, Lindquist D, et al. Lapatinib plus capecitabine for HER2-positive advanced breast cancer. N Engl J Med 2006; 355:2733–43.
- 11. Catalano V, Labianca R, Beretta GD, et al. Gastric cancer. Crit Rev Oncol Hematol 2005; 54:209–41.
- 12. Faivre J, Forman D, Esteve J, et al. Survival of patients with oesophageal and gastric cancers in Europe. Eur J Cancer 1998; 34:2167–75.
- 13. Power DG, Kelsen DP, Shah MA. Power Advanced gastric cancer--slow but steady progress. Cancer Treat Rev 2010; 36:384–92.

- 14. De Vivo R, Pignata S, Palaia R, et al. The role of chemotherapy in the management of gastric cancer. J Clin Gastroenterol 2000; 30:364–71.
- 15. Hofmann M, Stoss O, Shi D, et al. Assessment of a HER2 scoring system for gastric cancer: results from a validation study. Histopathology 2008; 52:797–805.
- Tanner M, Hollmen M, Junttila TT, et al. Amplification of HER2 in gastric cancer—association with topoisomerase IIa gene amplification, intestinal type, poor prognosis and sensitivity to trastuzumab. Ann Oncol 2005; 16:273–8.
- 17. Yoon HH, Shi Q, Sukov WR, et al. Association of HER2/ErbB2 expression and gene amplification with pathologic features and prognosis in esophageal adenocarcinomas. Clin Cancer Res 2012; 18:546–54.
- 18. Bang YJ, van Cutsem E, Feyereislova A, et al. Trastuzumab in combination with chemotherapy *versus* chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet 2010;376:687–97.
- 19. Albarello L, Pecciarini L, Doglioni C. HER2 testing in gastric cancer. Adv Anat Pathol 2011;18:53–9.
- 20. Junttila TT, Li G, Parsons K, et al. Trastuzumab-DM1 (T-DM1) retains all the mechanisms of action of trastuzumab and efficiently inhibits growth of lapatinib insensitive breast cancer. Breast Cancer Res Treat 2011; 128:347–56.
- 21. Issell BF, Crooke ST. Maytansine. Cancer Treat Rev 1978; 5:199–207.
- 22. Cassady JM, Chan KK, Floss HG, et al. Recent developments in the maytansinoid antitumor agents. Chem Pharm Bull (Tokyo) 2004; 52:1–26.
- 23. Cabanillas F, Chan KK, Floss HG, et al. Results of a Phase II study of maytansine in patients with breast carcinoma and melanoma. Cancer Treat Rep 1979; 63:507–9.
- 24. Erickson HK, Park PU, Widdison WC, et al. Antibody-maytansinoid conjugates are activated in targeted cancer cells by lysosomal degradation and linker-dependent intracellular processing. Cancer Res 2006; 66:4426–33.
- 25. Shen B-Q, Bumbaca D, Saad O, et al. Metabolic fate and pharmacokinetic characterization of trastuzumab emtansine (T-DM1): An emphasis on preclinical and clinical catabolism. ASCPT 2011.
- 26. Hurvitz SA, Dirix L, Kocsis J, et al. Phase II randomized study of trastuzumab emtansine versus trastuzumab plus docetaxel in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer. J Clin Oncol 2013;31(9):1157–63.
- 27. Verma S, Miles D, Gianni L, et al. Trastuzumab emtansine for HER2-positive advanced breast cancer. N Engl J Med 2012;367:1783–91.

- 28. Krop IE, Kim SB, González-Martín A, et al. Trastuzumab emtansine versus treatment of physician's choice for pretreated HER2-positive advanced breast cancer (TH3RESA): a randomised, open-label, phase 3 trial. Lancet Oncol 2014;15(7):689–99.
- 29. Beeram M, Krop IE, Burris HA, et al. A phase 1 study of weekly dosing of trastuzumab emtansine (T-DM1) in patients with advanced human epidermal growth factor 2-positive breast cancer. Cancer 2012;118(23):5733–40.
- 30. Krop IE, Beeram M, Modi S, et al. Phase I study of trastuzumab-DM1, an HER2 antibody-drug conjugate, given every three weeks to patients with HER2-positive metastatic breast cancer. J. Clin Oncol 2010; 28:2698–704.
- 31. Burris HA 3rd, Rugo HS, Vukelja SJ, et al. Phase II study of the antibody drug conjugate trastuzumab-DM1 for the treatment of human epidermal growth factor receptor 2 (HER2)-positive breast cancer after prior HER2-directed therapy. J Clin Oncol 2011;29(4):398–405.
- 32. Krop IE, LoRusso P, Miller KD, et al. A phase II study of trastuzumab emtansine in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer who were previously treated with trastuzumab, lapatinib, an anthracycline, a taxane, and capecitabine. J Clin Oncol 2012;30(26):3234–41.
- 33. Gupta M, Wang B, Carrothers TJ, et al. Effects of trastuzumab emtansine (T-DM1) on QT interval and safety of pertuzumab plus T-DM1 in patients with previously treated human epidermal growth factor receptor 2-positive metastatic breast cancer. Clinical Pharm in Drug Dev 2013;2:11–24.
- 34. Therasse P, Eisenhauer EA, Verwij J. RECIST revisited: a review of validation studies on tumour assessment. Eur J Cancer 2000; 42:1031–9.
- 35. Gupta M, LoRusso PM, Wang B, et al. Clinical implications of pathophysiological and demographic covariates on the population pharmacokinetics of trastuzumab-DM1, a HER2-targeted antibody–drug conjugate, in patients with HER2-positive metastatic breast cancer. J Clin Pharmacol 2011; 52:691–703.
- 36. Girish S, Gupta M, Wang B, et al. Clinical pharmacology of trastuzumab emtansine (T-DM1): an antibody–drug conjugate in development for the treatment of HER2-positive cancer. Cancer Chemother Pharmacol 2012; 69:1229–40.
- 37. Igawa Y, Matsubara M, Matsunaga K, et al. Pharmacokinetic (PK) and pharmacodynamic (PD) analysis of trastuzumab emtansine (T-DM1) in Japanese patients with advanced or recurrent HER2-positive breast cancer (JO22591): Comparison with Western patients. ASCPT 2012.
- 38. Blum JL, Dieras V, Lo Russo PM, et al. Multicenter, Phase II study of oral capecitabine in taxane-pretreated metastatic breast carcinoma patients. Cancer 2001; 92:1759–68.

- 39. Blum JL, Jones SE, Buzdar AU, et al. Multicenter Phase II study of capecitabine in paclitaxel-refractory metastatic breast cancer. J Clin Oncol 1999;17:485–93.
- 40. O'Shaughnessy , Miles D, Vukelja S, Moiseyenko V, Ayoub P, Cervantes G, Fumoleau P, Jones S, Lui WY, Mauriac L, Twelves C, Van Hazel G, Verma S, Leonard R. Superior survival with capecitabine plus docetaxel combination therapy in anthracycline-pretreated patients with advanced breast cancer: phase III trial results. J Clin Oncol 2002;20(12):2812–23.
- 41. Wardley A, Pivot X, Morales-Vasquez F, et al. Randomized phase II trial of first-line trastuzumab plus docetaxel and capecitabine compared with trastuzumab plus docetaxel in HER2-positive metastatic breast cancer. J Clin Oncol. 2010;28:976–83.
- 42. Sawaki A, Ohashi Y, Omuro Y, et al. Efficacy of trastuzumab in Japanese patients with HER2-positive advanced gastric or gastroesophageal junction cancer: a subgroup analysis of the Trastuzumab for Gastric Cancer (ToGA) study. Gastric Cancer 2012; 15:313–22.
- 43. Lewis Phillips G, Fields CT, Crocker L, et al. Potent anti-tumor activity of trastuzumab-DM1 antibody conjugate in combination with cytotoxic chemotherapeutic agents, antibodies or small molecule kinase inhibitors. AACR 2008; poster#2133.
- 44. Press MF, Sauter G, Bernstein L, et al. Diagnostic evaluation of HER-2 as a molecular target: an assessment of accuracy and reproducibility of laboratory testing in large, prospective, randomized clinical trials. Clin Cancer Res 2005; 11:6598–607.
- 45. Gelmon KA, Vidal M, Sablin M-P, et al. Trastuzumab emtansine (T-DM1) plus capecitabine (X) in patients with HER2-positive MBC: MO28230 TRAX-HER2 phase 1 results. J Clin Oncol 32:5s, 2014 (suppl; abstr 606).
- 46. Yang J, Wang Y, Zhao H, et al. Combination of exposure-response and case-control analyses in regulatory decision making. J Clin Oncol 2011; 29:(Suppl);4087.
- 47. Amstutz U, Froehlich TK, Largiadèr CR. Dihydropyrimidine dehydrogenase gene as a major predictor of severe 5-fluorouracil toxicity. Pharmacogenomics 2011;12(9):1321–36.
- 48. Drug Safety Report Xeloda and Fingerprint loss, 1067787, January 2016 (CDS Vs 14.0).

Trastuzumab Emtansine 598 RO5304020 Study MO28230

49. Moldoveanu Z, Huang W-Q, Kulhavy R, et al. Human male genital tract secretions: both mucosal and systemic immune compartments contribute to the humoral immunity. J Immunol 2005; 175:4127–36.

- 50. Rubinstein LV, Korn EL, Freidlin B, et al. Design issues of randomized phase II trials and a proposal for phase II screening trials. J Clin Oncol 2005;23:7199–206.
- 51. Ratain MJ, Sargent DJ. Optimising the design of phase II oncology trials: the importance of radnomisation. Eur J Cancer 2009;45:275–80.

Table 1 Schedule of assessments for mBC patients (Phase I, Cohort 1 and Randomized Phase II)

| Kadcy | | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | Сус | ele 4 Onw | ards | Safety<br>Follow-Up<br>Visit | Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Kadcyla (RO5304020) | Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 3-6<br>months |
| 040 | Informed Consent | Xa | | | | | | | | | | | |
| )20 | HER2 Status | Xp | | | | | | | | | | | |
| | Medical History and Demographics | X | | | | | | | | | | | |
| Roche | Complete Physical Examination | Х | | | | | | | | | | | |
| _ | Limited Physical Examination <sup>c</sup> | | Х | | | Х | | | Х | | | Х | |
| Clinical | Height and Weight <sup>d</sup> | Х | Х | | | Х | | | Х | | | Х | |
| al S | Vital Signs <sup>e</sup> | Х | Х | | | Х | | | Х | | | Х | |
| Study | ECOG Performance Status | Х | Х | | | Х | | | Х | | | Х | |
| | Concomitant Medication Reporting | X <sup>f</sup> | Х | | | | | Ongoir | ng | | | | |
| Report | AE Reporting | Xa | Ongoing | | | | | | | | Х | X <sup>h</sup> | |
| 1 | 12-lead ECG | Х | | | | | | | | | | | |
| Pro | ECHO/MUGA <sup>i</sup> | Xi | | | Xi | | | Xi | | | Xi | Xi | |
| Protocol MO28230 | Tumor Assessments <sup>j</sup> | х | At Cycle 3 (9 weeks after randomization), and then every 4 <sup>th</sup> cycle (12 weeks thereafter, regardless of dose delay or early discontinuation) until PD or study termination, X X whichever occurs earlier | | | | | | | | | | Х |
| )28 | Brain CT or MRI <sup>k</sup> | Х | | | At | the discre | etion of the | investiga | tor, if clinic | cally indica | ated, until F | -<br>PD | |
| 230 | Bone Scan/Imaging <sup>l</sup> | Х | | | | | , | As clinicall | y indicate | d | | | |

Kadcyla (RO5304020) Roche Clinical Study Report - Protocol MO28230 Research Report 1078906 1687

Appendix 1 Schedule of Assessments (cont.)

Schedule of assessments for mBC patients (Phase I, Cohort 1 and Randomized Phase II) (cont.) Table 1

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | Cycl | e 4 Onwa | rds | Safety<br>Follow-Up<br>Visit | Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 3-6<br>months |
| Hematology <sup>m</sup> | Х | Xn | Xn | Xn | Xn | Xn | Xn | Xn | | | Х | |
| Biochemistryº | X | Xn | Xn | Xn | Xn | Xn | Xn | Xn | | | Х | |
| Urinalysis <sup>p</sup> | X | | | | As clini | cally indic | ated | | | | Х | |
| INR/aPTT | Х | , | As clinically | indicated, | e.g. for pa | itients rec | eiving anti | coagulatio | n therapy | | Х | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Χq | | | Χq | Х | Х |
| PK Samples (see <u>Appendix 2</u> ) <sup>r</sup> | | Xr | | | Xr | | | | | | | |
| Assessment of Patient Hospitalizations and/or Hospital Visits | | х | | | Х | | | х | | | x | |
| Administration of Trastuzumab Emtansine | | D 2 <sup>s</sup> | | | D 1 <sup>s</sup> | | | D 1 <sup>s</sup> | | | | |
| Administration of Capecitabinet | | D. | 1–14 | | D 1 | <b>–14</b> | | D 1 | <b>–14</b> | | | |
| Overall Survival | | | | | | Х | | | | | Х | Х |
| Randomization into the Phase II Part of the Study | X <sup>ŧu</sup> | | | | | | | | | | | |

Research Report 1078906

# Appendix 1 Schedule of Assessments (cont.)

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

- 1.NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within **14 days** prior to first treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1).
- 2.All patients will be followed-up every 6 months (except for pregnancy, which is at 3 and 6 months after safety follow-up visit until disease progresses for tumor assessment or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than PD will continue to undergo tumor assessments every 3–6 months.
- a)Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests.
- b)HER2-positivity is defined as IHC 3+ or gene amplification by ISH. It will be performed locally for patients with mBC.
- c)Limited symptom-directed physical examination.
- d)Height to be obtained at screening or at Cycle 1 Day 1 only.
- e)Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f)Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to first study treatment.
- g)During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h)Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatment-related AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i)Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, between Days 15 and 21 in cycles 1 and 3, and between Days 15 and 21 of every third cycle thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

# Appendix 1 Schedule of Assessments (cont.)

- j)Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than PD, continued tumor assessments according to the protocol every 3–6 months until PD, withdrawal of consent, or study terminaton (whichever occurs earlier).
- k)Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 3 months) as detailed in Section 4.5.1.4 of the protocol and in Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- I)An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- m)Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and white blood cells (WBC) with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils.
- n)Assessments should be performed at screening, on Day 1, 8 and 15 of Cycles 1–3, on Day 1 of all subsequent cycles, and weekly following any hematologic AE. If capecitabine is discontinued due to toxicity, assessments should be performed weekly (minimum) until resolution of the AE (Grade ≤ 1/ baseline), and on Day 1 of subsequent cycles thereafter. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- o)Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, blood urea nitrogen (BUN)/urea (mandatory), creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN). Fasting is required before biochemistry assessment.
- p)Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.

# Research Report 1078906 1690

# Appendix 1 Schedule of Assessments (cont.)

- q)Serum β-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.
- r)Pharmacokinetic assessments will be performed during the MTD-Finding part of the study only (see Appendix 2).
- s)Trastuzumab emtansine will be administered on Day 1 of each 3-weekly cycle for all patients with mBC in Cohort 1 and Randomized Phase II period of the study except in the first cycle where trastuzumab emtansine will be given on Day 2 (to allow PK sampling).
- t) Capecitabine must be given within 30 minutes after a meal.
- u)Patients will be randomized only in the Randomized Phase II part of the study. No blinding will be used, as this is an open-label study.

# Kadcyla (RO5304020) Roche Clinical Study Report - Protocol MO28230 Research Report 1078906 1691

### Appendix 1 Schedule of Assessments (cont.)

Table 2 Schedule of assessments for patients with LA/mGC (Phase I, Cohort 2)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | Су | cle 4 Onw | ards | Safety<br>Follow-Up<br>Visit | Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28–42 days<br>after last<br>dose | every 3–6<br>months |
| Informed Consent | Xa | | | | | | | | | | | |
| HER2 Status | Xp | | | | | | | | | | | |
| Medical History and Demographics | Х | | | | | | | | | | | |
| Complete Physical Examination | Х | | | | | | | | | | | |
| Limited Physical Examination <sup>c</sup> | | Х | | | Х | | | Х | | | Х | |
| Height and Weight <sup>d</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Vital Signs <sup>e</sup> | Х | Х | | | Х | | | Х | | | Х | |
| ECOG Performance Status | Х | Х | | | Х | | | Х | | | Х | |
| Concomitant Medication Reporting | X <sup>f</sup> | Х | | | | | Ongoi | ng | | | | |
| AE Reporting | Xa | | | | | Ongoing | | | | | Х | X <sup>h</sup> |
| 12-lead ECG | Х | | | | | | | | | | | |
| ECHO/MUGA <sup>i</sup> | Xi | | | Xi | | | Xi | | | Xi | Xi | |
| Tumor Assessments <sup>j</sup> | Х | At 9 we | At 9 weeks after C1D1, and every 12 weeks thereafter, regardless of dose delay or early discontinuation, until PD or study termination, whichever occurs earliest | | | | | | | | | |
| Brain CT or MRI <sup>k</sup> | Х | | | Α | t the disc | retion of the | e investiga | tor, if clinic | cally indica | ated, until P | 'D | • |
| Bone Scan/Imaging <sup>l</sup> | Х | | | | | | As clinicall | y indicate | d | | | |

| Hematology <sup>m</sup> | Х | Xn | Xn | Xn | Xn | Xn | Xn | Xn | Xn | Xn | Х | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Biochemistryº | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | Xn | Xn | Xn | Xn | Xn | X <sup>n</sup> | Х | |
| Urinalysis <sup>p</sup> | Х | | | | As c | linically inc | dicated | | | | Х | |
| INR/aPTT | Х | P | s clinicall | y indicate | d, e.g. for | patients r | eceiving an | ticoagulat | ion therap | у | Х | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Χq | | | Xq | Х | Х |
| PK/PD Samples (see Appendix 2) | | Х | | | Х | | | | | | | |
| Assessment of Patient Hospitalizations and/or Hospital Visits | | Х | | | Х | | | Х | | | Х | |
| Administration of Trastuzumab Emtansine | | D 2 <sup>r</sup> | Х | Х | Х | х | х | Х | х | х | | |
| Administration of Capecitabines | | D 1- | -14 | | D 1 | -14 | | D 1 | -14 | | | |
| Overall Survival | | | | • | • | Х | • | • | | • | Х | Х |

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

Research Report 1078906

### Appendix 1 Schedule of Assessments (cont.)

- 1.NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within 14 days prior to first study treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1) visit.
- 2.All patients will be followed-up every 6 months (except for pregnancy, which is at 3 and 6 months after safety follow-up visit) until disease progresses for tumor assessment or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than PD will continue to undergo tumor assessments every 3-6 months.
- a)Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests.
- b)HER2-positivity is defined as IHC 3+ alone or IHC 2+ in combination with gene amplification by ISH. For patients with mGC enrolled into Cohort 2, central confirmation of HER2 status is required.
- c)Limited symptom-directed physical examination.
- d)Height to be obtained at screening or at Cycle 1 Day 1 only.
- e)Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f)Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to fist study treatment.
- g)During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h)Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatmentrelated AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i)Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, between Days 15 and 21 in cycles 1 and 3, and between Days 15 and 21 of every 3rd cycle thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

# Appendix 1 Schedule of Assessments (cont.)

- j)Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than PD, continue tumor assessments according to the protocol every 3–6 months until PD, withdrawal of consent, or study termination (whichever occurs earliest).
- k)Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 3 months) as detailed in Section 4.5.1.4 of the protocol and in Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- I)An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to first study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- m)Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and WBC with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils).
- n)Assessments should be performed at screening, on Day 1, 8 and 15 of all cycles. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- o)Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, BUN/urea (mandatory), creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN). Fasting is required before biochemistry assessment.
- p)Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.
- q)Serum β-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.
- r)Trastuzumab emtansine will be administered on Day 1 of each weekly cycle for all patients enrolled in Cohort 2 (A&B) except in the first cycle where trastuzumab emtansine will be given on DAY 2 (to allow drug interaction assessment).

s)Capecitabine must be given within 30 minutes after a meal.

# Appendix 2 Pharmacokinetic Sampling for Phase I, Metastatic Breast and Gastric Cancer Patients

| | Trastuzumab<br>emtansine, total<br>trastuzumab and DM1ª<br>PK samples (serum) | Capecitabine and 5-FU<br>PK samples (plasma) |
|---|---|---|
| Cycle 1 Day 1 | | |
| Pre-capecitabine dose | | Х |
| 30 min post capecitabine dosing | | X |
| 60 min post capecitabine dosing | | X |
| 1.5 hours post capecitabine dosing | | x |
| 2 hours post capecitabine dosing | | x |
| 2.5 hours post capecitabine dosing | | x |
| 4 hours post capecitabine dosing | | x |
| 6 hours post capecitabine dosing | | х |
| Cycle 1 Day 2 | | |
| Pre-trastuzumab emtansine dose | x | |
| 15-30 min after end of trastuzumab emtansine infusion | x | |
| Pre-capecitabine dose | | X |
| 30 min post capecitabine dosing | | X |
| 2 hours post capecitabine dosing | | x |
| 6 hours post capecitabine dosing | | x |
| Cycle 1 Day 3 | | |
| 24 hours (± 2 hours) after the end of infusion of trastuzumab emtansine | х | |
| Cycle 1 Day 9 | | |
| 7 days (± 1 day) after the end of infusion of trastuzumab emtansine <sup>a</sup> | х | |
| Cycle 2 Day 1 | | |
| Pre- capecitabine and trastuzumab emtansine dose <sup>a</sup> | x | |
| 15–30 min after end of trastuzumab emtansine infusion | x | |

### Trastuzumab emtansine—F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 4, 23 Mar 2016

| 30 min post capecitabine dosing | | х |
|---|---|---|
| 60 min post capecitabine dosing | | х |
| 1.5 hours post capecitabine dosing | | х |
| 2 hours post capecitabine dosing | | х |
| 2.5 hours post capecitabine dosing | | х |
| 4 hours post capecitabine dosing | | х |
| 6 hours post capecitabine dosing | | х |
| Cycle 2 Day 2 | | |
| 24 hours (± 2 hours) after the end of infusion of trastuzumab emtansine | x | |
| Cycle 2 Day 7 | | |
| 7 days (± 1 day) after the end of infusion of trastuzumab emtansine <sup>a</sup> | x | |
| Cycle 3 | | |
| Pre trastuzumab emtansine dose | x | |

PK = pharmacokinetic; 5-FU = 5-fluoruracil

Data from historic studies have determined that results are the lower limit of quantitation.

<sup>&</sup>lt;sup>a</sup> = Plasma DM1 samples will not be collected at Day 7 post-infusion of trastuzumab emtansine neither at pre-dose of Cycle 2 and Cycle 3.

Selected sections from the Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1,<sup>1</sup> are presented below, with slight modifications and the addition of explanatory text as needed for clarity.<sup>2</sup>

### Measurability of Tumor at Baseline

### **Definitions**

At baseline, tumor lesions/lymph nodes will be categorized as measurable or non-measurable as described below.

### a. Measurable Tumor Lesions

**Tumor Lesions.** Tumor lesions must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size as follows:

- 10 mm by CT or magnetic resonance imaging (MRI) scan (CT/MRI scan slice thickness/interval no greater than 5 mm)
- 10mm caliper measurement by clinical examination (lesions that cannot be accurately measured with calipers should be recorded as nonmeasurable)
- 20 mm by chest X-ray

**Malignant Lymph Nodes.** To be considered pathologically enlarged and measurable, a lymph node must be  $\geq$  15 mm in the short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and follow-up, only the short axis will be measured and followed. See also notes below on "Baseline Documentation of Target and Non-Target Lesions" for information on lymph node measurement.

<sup>&</sup>lt;sup>1</sup> Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (Version 1.1). Eur J Cancer 2009;45:228–47.

<sup>&</sup>lt;sup>2</sup> For consistency within this document, the section numbers and cross-references to other sections within the article have been deleted and minor formatting changes have been made.

### b. Non-Measurable Tumor Lesions

Non-measurable tumor lesions encompass small lesions (longest diameter > 10 mm or pathological lymph nodes with short axis ≥ 10 but < 15 mm) as well as truly non-measurable lesions. Lesions considered truly non-measurable include leptomeningeal disease, ascites, pleural or pericardial effusion, inflammatory breast disease, lymphangitic involvement of skin or lung, peritoneal spread, and abdominal mass/abdominal organomegaly identified by physical examination that is not measurable by reproducible imaging techniques.

### c. Special Considerations Regarding Lesion Measurability

Bone lesions, cystic lesions, and lesions previously treated with local therapy require particular comment, as outlined below.

### Bone Lesions:

- Bone scan, PET scan, or plain films are not considered adequate imaging techniques for measuring bone lesions. However, these techniques can be used to confirm the presence or disappearance of bone lesions.
- Lytic bone lesions or mixed lytic-blastic lesions, with identifiable soft tissue components, that can be evaluated by cross-sectional imaging techniques such as CT or MRI can be considered as measurable lesions if the soft tissue component meets the definition of measurability described above.
- Blastic bone lesions are non-measurable.

### Cystic Lesions:

- Lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor non-measurable) since they are, by definition, simple cysts.
- Cystic lesions thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of measurability described above. However, if non-cystic lesions are present in the same patient, these are preferred for selection as target lesions.

### Lesions with Prior Local Treatment:

 Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion. Study protocols should detail the conditions under which such lesions would be considered measurable.

### **Target Lesions: Specifications by Methods of Measurements**

### a. Measurement of Lesions

All measurements should be recorded in metric notation, using calipers if clinically assessed. All baseline evaluations should be performed as close as possible to the treatment start and never more than 28 days before the beginning of the treatment.

### b. Method of Assessment

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during the study. Imaging-based evaluation should always be the preferred option.

**Clinical Lesions.** Clinical lesions will only be considered measurable when they are superficial and ≥ 10 mm in diameter as assessed using calipers (e.g., skin nodules). For the case of skin lesions, documentation by color photography including a ruler to estimate the size of the lesion is suggested.

**Chest X-Ray.** Chest CT is preferred over chest X-ray, particularly when progression is an important endpoint, since CT is more sensitive than X-ray, particularly in identifying new lesions. However, lesions on chest X-ray may be considered measurable if they are clearly defined and surrounded by aerated lung.

**CT, MRI.** CT is the best currently available and reproducible method to measure lesions selected for response assessment. This guideline has defined measurability of lesions on CT scan based on the assumption that CT slice thickness is 5 mm or less. When CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness. MRI is also acceptable.

If prior to enrollment it is known that a patient is unable to undergo CT scans with IV contrast because of allergy or renal insufficiency, the decision as to whether a non-contrast CT or MRI (without IV contrast) will be used to evaluate the patient at baseline and during the study should be guided by the tumor type under investigation and the anatomic location of the disease. For patients who develop contraindications to contrast after baseline contrast CT is done, the decision as to whether non-contrast CT or MRI (enhanced or non-enhanced) will be performed should also be based on the tumor type and the anatomic location of the disease, and should be optimized to allow for comparison with the prior studies if possible. Each case should be discussed with the radiologist to determine if substitution of these other approaches is possible and, if not, the patient should be considered not evaluable from that point forward. Care must

be taken in measurement of target lesions on a different modality and interpretation of non-target disease or new lesions, since the same lesion may appear to have a different size using a new modality.

**Ultrasound.** Ultrasound is not useful in assessment of lesion size and should not be used as a method of measurement.

**Endoscopy, Laparoscopy, Tumor Markers, Cytology, Histology.** The utilization of these techniques for objective tumor evaluation cannot generally be advised.

### **Tumor Response Evaluation**

### Assessment of Overall Tumor Burden and Measurable Disease

To assess objective response or future progression, it is necessary to estimate the overall tumor burden at baseline and use this as a comparator for subsequent measurements. Measurable disease is defined by the presence of at least one measurable lesion, as detailed above.

### **Baseline Documentation of Target and Non-Target Lesions**

When more than one measurable lesion is present at baseline, all lesions up to a maximum of five lesions total (and a maximum of two lesions per organ) representative of all involved organs should be identified as target lesions and will be recorded and measured at baseline. This means that, for instances in which patients have only one or two organ sites involved, a maximum of two lesions (one site) and four lesions (two sites), respectively, will be recorded. Other lesions (albeit measurable) in those organs will be recorded as non-measurable lesions (even if the size is > 10 mm by CT scan).

Target lesions should be selected on the basis of their size (lesions with the longest diameter) and be representative of all involved organs, but in addition should lend themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion does not lend itself to reproducible measurement, in which circumstance the next largest lesion that can be measured reproducibly should be selected.

Lymph nodes merit special mention since they are normal anatomical structures that may be visible by imaging even if not involved by tumor. As noted above, pathological nodes that are defined as measurable and may be identified as target lesions must meet the criterion of a short axis of  $\geq 15$  mm by CT scan. Only the short axis of these nodes will contribute to the baseline sum. The short axis of the node is the diameter normally used by radiologists

to judge if a node is involved by solid tumor. Nodal size is normally reported as two dimensions in the plane in which the image is obtained (for CT this is almost always the axial plane; for MRI the plane of acquisition may be axial, sagittal, or coronal). The smaller of these measures is the short axis. For example, an abdominal node that is reported as being 20 mm × 30 mm has a short axis of 20 mm and qualifies as a malignant, measurable node. In this example, 20 mm should be recorded as the node measurement. All other pathological nodes (those with short axis ≥ 10 mm but < 15 mm) should be considered non-target lesions. Nodes that have a short axis of < 10 mm are considered non-pathological and should not be recorded or followed.

A sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the baseline sum of diameters. If lymph nodes are to be included in the sum, then, as noted above, only the short axis is added into the sum. The baseline sum of diameters will be used as a reference to further characterize any objective tumor regression in the measurable dimension of the disease.

All other lesions (or sites of disease), including pathological lymph nodes, should be identified as non-target lesions and should also be recorded at baseline. Measurements are not required and these lesions should be followed as "present," "absent," or in rare cases "unequivocal progression."

In addition, it is possible to record multiple non-target lesions involving the same organ as a single item on the Case Report Form (CRF) (e.g., "multiple enlarged pelvic lymph nodes" or "multiple liver metastases").

### **Response Criteria**

### a. Evaluation of Target Lesions

This section provides the definitions of the criteria used to determine objective tumor response for target lesions.

- Complete response (CR): Disappearance of all target lesions
   Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.</li>
- Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters
- Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline

In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.

The appearance of one or more new lesions is also considered progression.

 Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study

### b. Special Notes on the Assessment of Target Lesions

**Lymph Nodes.** Lymph nodes identified as target lesions should always have the actual short axis measurement recorded (measured in the same anatomical plane as the baseline examination), even if the nodes regress to < 10 mm on study. This means that when lymph nodes are included as target lesions, the sum of lesions may not be zero even if CR criteria are met, since a normal lymph node is defined as having a short axis of < 10 mm.

Target Lesions That Become Too Small to Measure. During the study, all lesions (nodal and non-nodal) recorded at baseline should have their actual measurements recorded at each subsequent evaluation, even when very small (e.g., 2 mm). However, sometimes lesions or lymph nodes that are recorded as target lesions at baseline become so faint on CT scan that the radiologist may not feel comfortable assigning an exact measure and may report them as being too small to measure. When this occurs, it is important that a value be recorded on the CRF, as follows:

- If it is the opinion of the radiologist that the lesion has likely disappeared, the measurement should be recorded as 0 mm.
- If the lesion is believed to be present and is faintly seen but too small to measure, a default value of 5 mm should be assigned and below measurable limit (BML) should be ticked. (Note: It is less likely that this rule will be used for lymph nodes since they usually have a definable size when normal and are frequently surrounded by fat such as in the retroperitoneum; however, if a lymph node is believed to be present and is faintly seen but too small to measure, a default value of 5 mm should be assigned in this circumstance as well and BML should also be ticked).

To reiterate, however, if the radiologist is able to provide an actual measure, that should be recorded, even if it is below 5 mm, and in that case BML should not be ticked.

**Lesions That Split or Coalesce on Treatment.** When non-nodal lesions fragment, the longest diameters of the fragmented portions should be added

together to calculate the target lesion sum. Similarly, as lesions coalesce, a plane between them may be maintained that would aid in obtaining maximal diameter measurements of each individual lesion. If the lesions have truly coalesced such that they are no longer separable, the vector of the longest diameter in this instance should be the maximum longest diameter for the coalesced lesion.

### c. Evaluation of Non-Target Lesions

This section provides the definitions of the criteria used to determine the tumor response for the group of non-target lesions. While some non-target lesions may actually be measurable, they need not be measured and instead should be assessed only qualitatively at the time points specified in the protocol.

- Complete response (CR): Disappearance of all non-target lesions and (if applicable) normalization of tumor marker level
  - All lymph nodes must be non-pathological in size (< 10 mm short axis).
- Non-CR/Non-PD: Persistence of one or more non-target lesions and/or (if applicable) maintenance of tumor marker level above the normal limits
- Progressive disease (PD): Unequivocal progression of existing non-target lesions

The appearance of one or more new lesions is also considered progression.

### d. Special Notes on Assessment of Progression of Non-Target Disease

When the Patient Also Has Measurable Disease. In this setting, to achieve unequivocal progression on the basis of the non-target disease, there must be an overall level of substantial worsening in non-target disease in a magnitude that, even in the presence of SD or PR in target disease, the overall tumor burden has increased sufficiently to merit discontinuation of therapy. A modest increase in the size of one or more non-target lesions is usually not sufficient to qualify for unequivocal progression status. The designation of overall progression solely on the basis of change in non-target disease in the face of SD or PR of target disease will therefore be extremely rare.

When the Patient Has Only Non-Measurable Disease. This circumstance arises in some Phase III trials when it is not a criterion of study entry to have measurable disease. The same general concepts apply here as noted above; however, in this instance there is no measurable disease assessment to factor into the interpretation of an increase in non-measurable disease burden. Because worsening in non-target disease cannot be easily quantified (by definition: if all lesions are truly non-measurable), a useful test that can be

applied when assessing patients for unequivocal progression is to consider if the increase in overall disease burden based on the change in non-measurable disease is comparable in magnitude to the increase that would be required to declare PD for measurable disease, that is, an increase in tumor burden representing an additional 73% increase in volume (which is equivalent to a 20% increase in diameter in a measurable lesion). Examples include an increase in a pleural effusion from "trace" to "large" or an increase in lymphangitic disease from localized to widespread, or may be described in protocols as "sufficient to require a change in therapy." If unequivocal progression is seen, the patient should be considered to have had overall PD at that point. While it would be ideal to have objective criteria to apply to non-measurable disease, the very nature of that disease makes it impossible to do so; therefore, the increase must be substantial.

### e. New Lesions

The appearance of new malignant lesions denotes PD; therefore, some comments on detection of new lesions are important. There are no specific criteria for the identification of new radiographic lesions; however, the finding of a new lesion should be unequivocal, that is, not attributable to differences in scanning technique, change in imaging modality, or findings thought to represent something other than tumor (e.g., some "new" bone lesions may be simply healing or flare of pre-existing lesions). This is particularly important when the patient's baseline lesions show partial or CR. For example, necrosis of a liver lesion may be reported on a CT scan report as a "new" cystic lesion, which it is not.

A lesion identified during the study in an anatomical location that was not scanned at baseline is considered a new lesion and will indicate PD.

If a new lesion is equivocal, e.g., because of its small size, continued therapy and follow-up evaluation will clarify if it represents truly new disease. If repeat scans confirm there is definitely a new lesion, then progression should be declared using the date of the initial scan.

### **Evaluation of Response**

### a. Time Point Response (Overall Response)

It is assumed that at each protocol-specified time point, a response assessment occurs. **Table 1** provides a summary of the overall response status calculation at each time point for patients who have measurable disease at baseline.

When patients have non-measurable (therefore non-target) disease only, **Table 2** is to be used.

Table 1 Time Point Response: Patients with Target Lesions (with or without Non-Target Lesions)

| Target Lesions | Non-Target Lesions | New Lesions | Overall Response |
|---|---|---|---|
| | CR | No | CR |
| CR | | | |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | NE |
| PD | Any | Yes or no | PD |
| Any | PD | Yes or no | PD |
| Any | Any | Yes | PD |

CR=complete response; NE=not evaluable; PD=progressive disease; PR=partial response; SD=stable disease.

Table 2 Time Point Response: Patients with Non-Target Lesions Only

| Non-Target Lesions | New Lesions | Overall Response |
|--------------------|-------------|----------------------------|
| | No | CR |
| CR | | |
| Non-CR/non-PD | No | Non-CR/non-PD <sup>a</sup> |
| Not all evaluated | No | NE |
| Unequivocal PD | Yes or no | PD |
| Any | Yes | PD |

 $\label{eq:crossing} \mbox{CR=complete response; NE=not evaluable; PD=progressive disease.}$ 

a "Non-CR/non-PD" is preferred over "stable disease" for non-target disease since stable disease is increasingly used as an endpoint for assessment of efficacy in some trials; thus, assigning "stable disease" when no lesions can be measured is not advised.

### b. Missing Assessments and Not Evaluable Designation

When no imaging/measurement is done at all at a particular time point, the patient is not evaluable at that time point. If only a subset of lesion measurements are made at an assessment, usually the case is also considered not evaluable at that time point, unless a convincing argument can be made that the contribution of the individual missing lesion(s) would not change the assigned time point response. This would be most likely to happen in the case of PD. For example, if a patient had a baseline sum of 50 mm with three measured lesions and during the study only two lesions were assessed, but those gave a sum of 80 mm, the patient will have achieved PD status, regardless of the contribution of the missing lesion.

If one or more target lesions were not assessed either because the scan was not done or the scan could not be assessed because of poor image quality or obstructed view, the response for target lesions should be "unable to assess" since the patient is not evaluable. Similarly, if one or more non-target lesions are not assessed, the response for non-target lesions should be "unable to assess" except where there is clear progression. Overall response would be "unable to assess" if either the target response or the non-target response is "unable to assess" except where this is clear evidence of progression, as this equates with the case being not evaluable at that time point.

### c. Special Notes on Response Assessment

When nodal disease is included in the sum of target lesions and the nodes decrease to "normal" size (<10 mm), they may still have a measurement reported on scans. This measurement should be recorded even though the nodes are normal in order not to overstate progression should it be based on increase in size of the nodes. As noted earlier, this means that patients with CR may not have a total sum of "zero" on the CRF.

Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of PD at that time should be reported as "symptomatic deterioration." Every effort should be made to document objective progression even after discontinuation of treatment. Symptomatic deterioration is not a descriptor of an objective response; it is a reason for stopping study therapy. The objective response status of such patients is to be determined by evaluation of target and non-target disease as shown in **Table 1**, **Table 2**, **Table 3**.

Table 3 Best Overall Response When Confirmation Is Required

| Overall Response at First Time Point | Overall Response at<br>Subsequent Time Point | Best Overall Response |
|---|---|---|
| | CR | CR |
| CR | | |
| CR | PR | SD, PD, or PR <sup>a</sup> |
| CR | SD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| CR | PD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| CR | NE | SD, provided minimum<br>duration for SD was met;<br>otherwise, NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | SD, provided minimum<br>duration for SD was met;<br>otherwise, PD |
| PR | NE | SD, provided minimum<br>duration for SD was met;<br>otherwise, NE |
| NE | NE | NE |

CR=complete response; NE=not evaluable; PD=progressive disease; PR=partial response; SD=stable disease

<sup>&</sup>lt;sup>a</sup> If a CR is truly met at the first time point, any disease seen at a subsequent time point, even disease meeting PR criteria relative to baseline, qualifies as PD at that point (since disease must have reappeared after CR). Best response would depend on whether the minimum duration for SD was met. However, sometimes CR may be claimed when subsequent scans suggest small lesions were likely still present and in fact the patient had PR, not CR, at the first time point. Under these circumstances, the original CR should be changed to PR and the best response is PR.

For equivocal findings of progression (e.g., very small and uncertain new lesions; cystic changes or necrosis in existing lesions), treatment may continue until the next scheduled assessment. If at the next scheduled assessment, progression is confirmed, the date of progression should be the earlier date when progression was suspected.

In studies for which patients with advanced disease are eligible (i.e., primary disease still or partially present), the primary tumor should also be captured as a target or non-target lesion, as appropriate. This is to avoid an incorrect assessment of CR if the primary tumor is still present but not evaluated as a target or non-target lesion.

# Appendix 4 Instructions for Scans in the Event of Isotope Shortage

Two key suppliers of Tc-99m generators (Chalk River Reactor, Canada and High Flux Reactor, the Netherlands) are expected to close. Supplies from other reactor sources will be unable to meet the expected world-wide patient-care needs. As a result, significant shortages of Tc-99m are expected, and the instructions listed below should be followed:

- ECHO will be the preferred imaging modality over MUGA scans to evaluate cardiac function.
- Tc-99m bone scans should be obtained as part of the baseline tumor assessment in all patients and should be repeated to confirm a CR or if progression of existing bone lesions and/or the development of new bone lesions is clinically suspected.
  - If a bone scan cannot be performed at baseline or if the investigator suspects that a bone scan may not be able to be repeated during the course of the study because of the Tc-99m shortage, the investigator may choose F-18 NaF or FDG-PET scan as an alternative.
- If bone lesions are selected as index non-target lesions, they must be apparent on baseline CT scans or other radiographic modalities (e.g., skeletal X-rays that can be repeated in subsequent tumor assessments). Additional scans may be obtained to follow clinically important bone lesions if not visualized on the chest, abdomen, or pelvic CT scan.

These measures are intended to ensure that the same method of assessment and the same imaging technique is used throughout the study for each patient. If there is a question regarding the choice of alternatives in the event that a standard bone scan cannot be obtained during screening and/or during the study, please contact the Medical Monitor.

# Appendix 5 New York Heart Association Classification of Functional Cardiac Capacity

| Class | |
|---|---|
| I | No limitation: Ordinary physical activity does not cause undue fatigue, dyspnea, or palpitation. |
| II | Slight limitation of physical activity: Such patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitations, dyspnea, or angina. |
| III | Marked limitation of physical activity: Although patients are comfortable at rest, less than ordinary physical activity will lead to symptoms. |
| IV | Inability to carry on physical activity without discomfort: Symptoms of congestive heart failure are present even at rest. With any physical activity, increased discomfort is experienced. |

From: Criteria Committee, New York Heart Association, Inc. Diseases of the heart and blood vessels. Nomenclature and criteria for diagnosis. 6th ed. Boston, Little, Brown and Co, 1964:114.
# Appendix 6 ECOG Performance Status

| | Scale |
|---|---|
| Grade | |
| 0 | Fully active able to carry on all pre-disease performance |
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, |
| 2 | i.e., light housework, office work Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair |
| 5 | Dead |

52. http://www.ecog.org/general/perf\_stat.html

#### **PROTOCOL**

TITLE: PHASE I STUDY OF THE COMBINATION OF

TRASTUZUMAB EMTANSINE (T-DM1) AND

CAPECITABINE IN HER2-POSITIVE METASTATIC
BREAST CANCER AND HER2-POSITIVE LOCALLY
ADVANCED OR METASTATIC GASTRIC CANCER
PATIENTS, FOLLOWED BY A RANDOMIZED,
OPEN-LABEL PHASE II STUDY OF T-DM1 AND
CAPECITABINE VERSUS T-DM1 ALONE IN HER2POSITIVE METASTATIC BREAST CANCER

PROTOCOL NUMBER: MO28230

**EUDRACT NUMBER:** 2012-001547-46


MEDICAL MONITOR: MD

**SPONSOR:** F. Hoffmann-La Roche Ltd

**DATE FINAL:** Version : 21-Aug-2012

**DATE AMENDED:** Version: 03-Sep-2013

### PROTOCOL AMENDMENT APPROVAL

## **CONFIDENTIAL STATEMENT**

The information contained in this document, especially any unpublished data, is the property of F. Hoffmann-La Roche Ltd (or under its control) and therefore is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Ethics Committee or Institutional Review Board. It is understood that this information will not be disclosed to others without written authorization from Roche except to the extent necessary to obtain informed consent from persons to whom the drug may be administered.

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd Protocol MO28230, Version 2, 03 September 2013

# PROTOCOL AMENDMENT, VERSION 2 RATIONALE

Roche is performing continuous characterization of the trastuzumab emtansine (T-DM1) safety profile to ensure patient safety is maintained.

The recently released Investigator Brochure (IB) version 7.0 includes recent safety and clinical data analyses leading to updated guidance on dose modification. This dose modification guidance is now reflected in this protocol amendment. As stated in the IB v.7.0, these updates have no impact on the overall assessment of risk and benefit with T-DM1.

To date, a total of seven patients have been treated at the dose level 750 mg/m² capecitabine. Two dose-limiting toxicities (DLTs), one case of nausea and vomiting and one case of a Grade 3 alanine transaminase (ALT) elevation, were observed in two patients in this cohort. Both DLTs prevented Cycle 2 restarting at 100% of the dose on Cycle 2 Day 1. Another patient in this cohort showed ALT and aspartate transaminase (AST) elevation without meeting the DLT criteria. A retrospective eligibility review showed that this patient had not fulfilled completely the IB requirement of stable liver function tests prior to study enrollment. Although the patient did not meet the DLT criteria as per protocol, the patient was replaced by a 7<sup>th</sup> patient, following the Steering Committee (SC) recommendation, to ensure that another, more informative patient was included to avoid any bias while evaluating the drug effect. Following the investigator assessment and the SC recommendation, we believe, as a Sponsor, that the available evidence shows an acceptable positive risk-benefit in all seven patients treated at Dose Level 1.

As of 7 August 2013, five patients remain on treatment, with a follow-up period of 4 to 8 months. Of the two patients who have discontinued treatment, one patient's disease has progressed, and the other discontinuation was based on the investigator's decision, following the central confirmation, that the patient's disease was HER2-negative. Considering the available safety data for all patients (maximum number of cycles is 12), the combination of capecitabine and T-DM1 is well tolerated, except for increases in transaminases and hand-foot syndrome. Dose modifications of T-DM1 and/or capecitabine have allowed those patients to continue on treatment. No serious adverse events have been reported and responses have been observed in six patients. Latest tumor response data show two patients with partial response (PR) and four patients with stable disease (SD). In view of the two DLT events in Cohort 1, the SC has recommended the combination of T-DM1 and capecitabine to be further explored by introducing a lower-dose cohort of capecitabine.

This protocol amendment aims to further clarify patient retention on combination regimen. This will allow an additional safety follow-up and collection of tumor response from these patients on combination treatment whilst the SC and the Sponsor continually monitor the risk-benefit profile of the combination treatment.

The design of the Phase II part of the study has been changed to the openlabel, randomized Phase II study to explore the efficacy and safety of the combination of T-DM1 with capecitabine compared with T-DM1 alone. A 2:1 randomization was chosen to allow more patients being exposed to the combination of T-DM1 and capecitabine. This will enable a more thorough assessment of the corresponding safety profile.

1. Changes according to IB v.7.0.

The following sections were updated with the latest clinical information and current recommendations:

- 5.1.1 Risks associated with trastuzumab emtansine (including thrombocytopenia, hepatotoxicity, infusion-related reactions/hypersensitivity, pulmonary toxicity, neurotoxicity, cardiotoxicity, and extravasation)
- 5.1.2 Risks associated with capecitabine (including cardiotoxicity, DPD deficiency, hand-foot syndrome, and hepatotoxicity)
- 5.1.3 Trastuzumab emtansine and capecitabine combination
- 5.1.4 Definition of the dose limiting toxicity
- 5.1.5.1 Trastuzumab emtansine dose modification (including dose modification for thrombocytopenia, hepatotoxicity, neurotoxicity, cardiotoxicity, infusion-related reactions, hypersensitivity reactions, pulmonary toxicity, and extravasation)
- 5.1.5.2 Capecitabine dosage modification
- 2. Changes for introducing lower doses of capecitabine.
  - Dose Levels -1 (700 mg/m²) and -2 (650 mg/m²) have been added
  - Rules for escalation and de-escalation of capecitabine doses have been amended to allow de-escalation from Dose Level 1 to Dose Levels -1 and -2 in case of toxicity. No re-escalation to Dose Level 1 is allowed
  - The doses of 750 mg/m<sup>2</sup> and higher will not be further explored
  - The DLT criteria will not be changed, but the SC adjudication will be permitted in cases not covered by the criteria
  - Patients who are currently receiving capecitabine 750 mg/m<sup>2</sup> can continue with the dose
- 3. Changes for introducing the open-label, Randomized Phase II part of the study instead of Cohort 1, Phase II
  - Protocol title has been amended to reflect the change in study design
  - Objectives of the Phase II part of the study has been amended to include new treatment groups
  - Sample size for Phase II has been recalculated based on estimated best overall response (BOR) for the combination treatment and T-DM1 alone
  - Number of patients in Phase II and in the whole study has been amended according to the new sample size calculation

- A medical justification has been added for the estimation of BOR for the combination treatment
- Independent Data Monitoring Committee (IDMC) for Phase II has been introduced to monitor safety outcomes
- 4. Changes for protocol consistency.
  - The Protocol (Amendment) Acceptance Form has been updated according to the latest approved wording

Additional minor changes have been made to improve clarity and consistency. Deleted text appears in red strikethrough. Substantive new information is marked with yellow highlighting. This amendment represents cumulative changes to the original protocol.

# PROTOCOL AMENDMENT, VERSION 2 SUMMARY OF CHANGES

## **TITLE PAGE**

TITLE: PHASE I FOLLOWED BY PHASE II STUDY OF THE

COMBINATION OF TRASTUZUMAB EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED OR METASTATIC GASTRIC CANCER PATIENTS, FOLLOWED BY A RANDOMIZED, OPEN-LABEL PHASE II STUDY OF T-DM1 AND CAPECITABINE VERSUS T-DM1 ALONE IN HER2-POSITIVE METASTATIC BREAST CANCER

## **SYNOPSIS**

#### **Objectives**

Randomized Phase II: Exploration of Efficacy and Safety in mBC

Primary Objective:

- ORR by investigator assessment
- To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine in mBC patients, as measured by ORR by Response Evaluation Criteria for Solid Tumors (RECIST) v.1.1 per investigator local assessment

#### Secondary Objectives

- Safety profile of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine
- To explore the dose established during Phase lefficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine in mBC patients, as measured by:

## Study Design

#### **Description of Study**

This is an international, multicenter study.

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in human epidermal growth factor receptor 2 (HER2)-positive mBC and locally advanced or mGC patients, using a Phase I design, followed by a randomized, open-label Phase II-single arm study to explore the efficacy and safety of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine in mBC patients. There will be no exploration of efficacy in the mGC cohort. Results from the Phase I in mGC will be used as supporting information for future studies in the indication (see Figure 4 in the protocol).

Cohort 1 (mBC) and Cohort 2 (mGC) will open sequentially during Phase I.

#### Phase I: MTD Finding, Cohort 1: mBC

Cohort 1 will open first with a 3 plus 3 classical design. Cohort 1 will enroll patients with HER2-positive mBC. The dose tested of trastuzumab emtansine remains fixed at 3.6 mg/kg every 3 weeks (q3w) and 3 dose levels of capecitabine administered twice daily (bid) on Days 1 to 14 in cycles of 3 weeks will be tested. All patients will be treated until disease progression, intolerable toxicity, withdrawn consent, or death. All patients will be followed-up intolerable toxicity, until withdrawn consent, death, or up to a maximum of 2 years after the last patient was enrolled randomized in the Phase II part of the study, whichever occurs first.

Dose Levels Explored in Phase I, Cohort 1

Dose Level 1: 750 mg/m² capecitabine twice daily (bid) + 3.6 mg/kg every three weeks (q3w) trastuzumab emtansine

# Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 42, 03 September 2013

Dose Level 2-1: 85700 mg/m² capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine Dose Level 3-2: 100650 mg/m² capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine The rules for dose escalation determining the MTD are presented below.

If Dose Level 1 is proved too toxic (dose-limiting toxicity [DLT] > 1/3 or > 1/6), the dose will be de-escalated to one dose level below (Dose Level -1)

If Dose Level -1 is well tolerated (DLT ≤ 1/6), this dose will be considered the MTD and, following the independent Data Monitoring Committee (IDMC) agreement, will be further explored in the Randomized Phase II part of the study. If Dose Level -1 is too toxic (DLT >1/6), the dose will be de-escalated to Dose Level -2.

If Dose Level -2 is well tolerated (DLT ≤ 1/6), this dose will be considered the MTD and, following iDMC approval, will be further explored in the Randomized Phase II part of the study. However, if Dose Level -2 is too toxic (DLT > 1/6), the combination may be considered unfeasible, recruitment will be closed and no other neither the Randomized Phase II nor mGC cohort will be opened. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the Steering Committee (SC).

Randomized Phase II: Exploration of Efficacy, Cohort 1: and Safety in mBC Phase II will be conducted in mBC patients only. This part of the study will explore the efficacy and safety of the combination treatment of T-DM1 and capecitabine, at the established MTD, compared with T-DM1 alone in mBC patients.

Once the MTD in Cohort—1 is established, recruitment into this cohort will be extended to a total of 110 additional 117 HER2-positive mBC patients forwill be randomized into the Phase II part of the study. Patients, who are on the MTD established in the Phase I part of the study, must re consent to be enrolled into Phase II. will not contribute to the Phase II part of the study; however, they will be followed-up until end of study (EOS).

Patients will be treated until disease progression/recurrence, intolerable toxicity, withdrawn consent, or death. If capecitabine needs to be discontinued for any reason, trastuzumab emtansine may continue, and the patient will remain evaluable in the study.be followed-up until EOS. In case of discontinuation of trastuzumab emtansine, patients will be withdrawn-from the study/followed-up until EOS.

All patients will be followed-up until disease progression, intolerable toxicity, withdrawn consent, death, or up to a maximum of 2 years after the last patient was enrolledrandomized in the Phase II part of the study, whichever occurs first. Patients who have not progressed at that point in time may be enrolled into an extension study.

#### Phase I: MTD Finding, Cohort 2: mGC

Once the capecitabine MTD dose is established in Cohort 1, Cohort 2 will open, with a 3 plus 3 classical design to enroll HER2-positive mGC patients. Trastuzumab emtansine will be administered weekly at the dose of 2.4 mg/kg and capecitabine will start at the MTD dose defined in Cohort 1; capecitabine dose level may be de-escalated.

All patients will be treated until disease progression, intolerable toxicity, withdrawn consent, or death. All patients will be followed-up until intolerable toxicity, withdrawn consent, death, or up to a maximum of 2 years after the last patient was enrolledrandomized in the Phase II part of the study, whichever occurs first.

The dose levels for capecitabine will be the same as described in Cohort 1, except for Dose Level 1, which will not be explored in mGC patients. Guidelines for dose escalation and descalation are as follows:

If the MTD established in Cohort 1 is defined at Dose Level 1 of 750 mg/m<sup>2</sup> bid-1:

- Escalation This will be tethe starting dose in Cohort 2. If Dose Level 2 of 850 mg/m² bid. 1 is well tolerated (DLT ≤ 1/6), this dose will be established as the MTD for mGC
- De-escalation: if Dose Level -1 is not tolerated (>1/3 or >in Cohort 2 (> 1/6 DLT), de-escalation will be to Dose Level -2

If the MTD established in Cohort 1 is defined at Dose Level -2:

 This will be the starting dose in Cohort 2. If Dose Level -2 is well tolerated (DLT ≤ 1/6), this dose will be established as the MTD for mGC De-escalation: if Dose Level -2 is not tolerated in Cohort 2 (> 1/6 DLT), the combination will be considered not feasible. for mGC and Cohort 2 will be terminated. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the SC

If MTD defined at Dose Level 2 of 850 mg/m<sup>2</sup> bid:

- Escalation will be to Dose Level 3 of 1000 mg/m<sup>2</sup> bid
- De escalation will be to Dose Level 1 of 750 mg/m<sup>2</sup> bid

If MTD defined at Dose Level 3 of 1000 mg/m<sup>2</sup> bid

- Escalation: There will be no escalation, MTD will be defined at Dose Level 3
- De escalation will be to Dose Level 2 of 850 mg/m<sup>2</sup> bid

#### **Number of Patients**

Phase I, Cohort 1: mBC

3A minimum of 6 and up to 18 patients maywill be enrolled.

Randomized Phase II: Exploration of Efficacy and Safety in mBC

Cohort 1 Exploration of efficacy and safety in mBC will be expanded to enroll 110 based on 117 randomized patients in total.

Phase I, Cohort 2: mGC

A total of 3 to 1812 patients maywill be enrolled.

#### **Target Population**

Phase I, Cohort 1: mBC

HER2-positive mBC patients will be enrolled.

The patient's HER2 status will be considered positive if the local institution or reference lab reported Grade 3+ staining intensity (on a scale of 0 to 3) by means of immunohistochemistry (IHC) or fluorescent *in situ* hybridization (FISH).

The HER2 status will be retrospectively confirmed by IHC and/or FISH in a central laboratory using archival paraffin-embedded tumor tissue. Patients must have received at least one metastatic disease and/or locally recurrent disease not amenable to resection. Retrospective central confirmation will not impact the treatment regimen decisions or primary endpoint of Phase I and will be used to validate efficacy analyses in Phase I.

Patients must have received at least one treatment regimen, which includes a chemotherapy agent and trastuzumab-agent.

Randomized Phase II, Cohort 1: Exploration of Efficacy and Safety in mBC

HER2-positive mBC patients will be enrolled randomized to one of the treatment groups receiving either the combination of trastuzumab emtansine (T-DM1) with capecitabine or T-DM1 alone. Retrospective central confirmation will be used to censor the efficacy population for the Randomized Phase II part of the study.

Patients must have received at least one treatment regimen, which includes a chemotherapy agent and trastuzumab-agent.

Phase I, Cohort 2: mGC

HER2-positive locally advanced or mGC patients will be enrolled.

Patients must not have received prior chemotherapy for advanced/metastatic disease.

Inclusion Criteria:

## For mBC Patients:

- 8. Liver function:
  - a) Total bilirubin ≤ 1.5 × the upper limit of normal (ULN), except in patients with previously documented Gilbert's syndrome in which case total bilirubin ≤ 3 mg/dLisacceptable
  - d) Evidence of stable liver function during the month prior to enrollment with liver function tests' (LFTs) fluctuations not exceeding 2.5 × ULN (for AST, ALT) and 1.5 × ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN.

14. mBC with at least one measurable lesion according to RECIST v.1.1.

#### For mGC Patients:

- 8. Liver function:
  - a) Total bilirubin ≤ 1.5 × ULN except in patients with previously documented—Gilbert's syndrome in which case total bilirubin ≤ 3 mg/dL is acceptable
  - d) Evidence of stable liver function during the month prior to enrollment with LFTs fluctuations not exceeding 2.5 × ULN (for AST, ALT) and 1.5 × ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN.
- 11. Histologically or cytologically confirmed GGmGC or locally advanced gastric cancer. Exclusion Criteria:

#### For mBC Patients:

- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product.
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 360500 mg/m<sup>2</sup>.
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 360500 mg/m² doxorubicin.
- 9. Current peripheral neuropathy of Grade ≥ 3 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v4.0.

#### For mGC Patients:

- 22. No signs and symptoms suggestive that the patient has DPD deficiency
- 23. Lapatinib ≤ 14 days before first study drug administration

#### Length of Study

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to be 2 years for Dose Finding and the Phase II/Exploration of Efficacy and Safety. All patients will be followed-up until intolerable toxicity, withdrawn consent, death or up to a maximum of 2 years after the last patient was enrolled randomized in the Phase II part of the study, whichever occurs first. In case Dose Level 4-2 is too toxic, the study may be terminated prematurely. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the SC.

#### **Efficacy Outcome Measures**

Efficacy will be evaluated as per RECIST v.1.1.

- · Best overall response (BOR) rate
- DoR
- TTR
- TTP
- TTF
- PFS
- CBR
- OS

#### **Safety Outcome Measures**

- DLT assessment
- Incidence and severity by NCI CTCAE version 4.0 of adverse events (AEs) and), serious adverse events (SAEs), AEs that cause discontinuation from the study treatment, and AEs of special interest (AESIs)
- CasesFatal cases and causes of death

#### **Pharmacokinetic Outcome Measures**

 PK will be evaluated during Phase I for both trastuzumab emtansine and capecitabine (see Appendix 1, Schedule of Assessment in the protocol). In addition, PK samples may be taken ad hoc, in case of SAE or unexpected toxicities, which may be suggestive of potential drug-drug interaction.

#### **Investigational Medicinal Products**

# Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 42, 03 September 2013

#### For mBC Patients:

<u>Capecitabine</u> will be administered twice a day, orally for 14 days followed by a 7-day rest period at the Dose Levels 1—3 to -2 described in the 'Trial Design' section.

Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Rounding of capecitabine dose, based on 150 mg and 500 mg tablet strength will be allowed to the nearest target dose, based on patient body surface area (BSA).

#### For mGC Patients:

<u>Capecitabine</u> will be administered twice a day, orally for 14 days followed by a 7-day rest period at the <u>dose levels 1 3Dose Levels -1 to -2</u> described in the 'Trial Design' section. Capecitabine tablets should be swallowed with water within 30 minutes after a meal.

#### Statistical Analysis

The study will include 2 phases and 2 cohorts:

- Phase I, Cohort 1: mBC Dose Finding Cohort
- Randomized Phase II, Cohort 1: mBC: Exploration of Efficacy Cohortand Safety in mBC
- Phase I, Cohort 2: mGC Dose Finding Cohort

During Phase I, the primary objective is reaching the MTD and establishing a safety profile.

There is no formal efficacy interim analysis. However, an independent data monitoring committee (IDMC) will advise whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 20 and 60 patients have received at least 3 cycles of treatment (Cycle 3 Day 1) in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II of the study or as requested.

Efficacy data will only be provided if required by the IDMC to estimate the risk-benefit balance for the patients. Further details on the function and logistics of the IDMC will be provided in the IDMC Charter.

Corresponding analyses as described in the protocol will be performed when all data for both cohorts and study phases are collected and cleaned.

#### Analysis of primary and secondary endpoints:

#### **Analysis Populations:**

Phase-I, Cohort 1: MTD Finding: mBC Patients:

The main analysis population will befor DLT assessment is the DLT evaluable population, which is defined as all enrolled and treated patients who have not experienced any major protocol violations (including violations of the inclusion and exclusion criteria) and have completed Cycle 1.

The safety population including(SP) will include all patients in this cohort who received at least one dose of study medication (trastuzumab emtansine and capecitabine) during this phase.

Phase I.

#### Randomized Phase II: Exploration of Efficacy: and Safety in mBC Patients

The main analysis population for the efficacy analysis will be the intent-to-treat (ITT) population-(ITT) including, which will include all new patients enrolled in Phase II and patients from Cohort 1 who achieved the MTD level randomized in the Phase II part of the study. The per-protocol (PP) population will include all ITT patients who have at least one post-baseline tumor assessment during the Phase-II II part of the study and no major protocol violations, which will be defined in the statistical analysis plan. Safety parameters-will be summarized for the safety population that includes all patients who received at least one dose of study medication in this part of the study. (SAP).

The SP will include all patients who received at least one dose of study medication during the Randomized Phase II part of the study.

## Phase I, Cohort 2: MTD Finding, mGC Patients:

The main analysis population will be for DLT assessment is the safety DLT evaluable population-, which is defined as all enrolled and treated patients who have not experienced any major protocol violation (including violation of the inclusion and exclusion criteria) and have completed Cycle 1.

Trastuzumab Emtansine—F. Hoffmann-La Roche Ltd Protocol MO28230, Version 42, 03 September 2013

The SP will include all patients in this cohort who received at least one dose of study medication (trastuzumab emtansine and capecitabine) during this phasePhase I.

#### Efficacy Endpoints:

#### Phase-I, Cohort 1: MTD Finding, mBC

The primary objectives are reaching the MTD and establishing a safety profile.

ORR, as a main efficacy endpoint, will be assessed via BORRBOR rate. The BOR is defined as the best response recorded from the date when the MTD is achieved of enrollment until disease progression/recurrence-(or, death)., withdrawal of consent or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### Randomized Phase\_II: Exploration of Efficacy: in mBC

The primary efficacy endpoint for the Phase—II part of the study is the BORORR, as assessed by investigaters via BOR. The BOR is defined as the best response recorded from the start of this or randomization into the Phase—III part of the study and until disease progression or recurrence (or, death) or for patients who were involved in Phase I of the study: the best response from the date, withdrawal of the MTD reached until disease progression/recurrence consent or death EOS, whichever occurs first. To be assigned a status of partial response (PR) or complete response (CR), i.e., to be a responder, changes in tumor measurements must be confirmed by repeatrepeated assessments that should be performed no less than 28 days after the response criteria for response are first met, i.e., patients need to have two consecutive assessments of PR or CR. This status will be assessed only for patients with measurable disease at baseline. Patients with non-measurable disease at baseline will be assessed for the time to event endpoints (e.g. PFS, OS, etc).

The emphasis of the exploratory Randomized Phase II part of the study will not be formal statistical hypothesis testing but the estimation of:

- The BOR rate with corresponding 95% confidence intervals (CIs) for each treatment group. The justification of the sample size is based on considerations regarding the width of 95% CIs for each treatment group estimate (precision of the corresponding estimate).
- The treatment effect (between treatment groups comparison) with corresponding 95% Cls.

The number and proportions of responders and non-responders (based on BOR) together with the two-sided, 95% Clopper-Pearson confidence intervals Cls will be presented. CBR-will be summarized for each treatment group. The difference in a similar way.BOR between treatment groups will be displayed with associated 95% Cls using the Hauck-Anderson approach.

The secondary endpoints for the Phase-II part of the study will be:

- Time to response (TTR)
- Duration of response (DoR)
- Time to progression (DoR)
- TTP)
- Time to treatment failure (TTF)
- Progression free survival (PFS)
- Clinical benefit rate (CBR)
- Overall survival (OS)
- TTF
- PFS
- CBR
- OS

Estimates for the survivor function for the time to event variable such as of both treatment groups for TTR, DoR, TTP, TTF, PFS, and OS, will be obtained by using the Kaplan-Meier approach, method. Hazard ratios and associated 95% CIs will be estimated from non-stratified and stratified (based on the stratification factor) Cox regression models.

Clinical benefit response will include patients whose best (confirmed) response was PR or CR, or stable disease (SD) that lasted at least 6 months. CBR will be summarized in a similar way to the primary efficacy endpoint, ORR, as assessed by BOR.

#### Safety Endpoints:

#### Phase-I, Cohort 1: MTD Finding: mBC

The number and proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

Safety parameters for this study part will be summarized by treatment dose. The summaries of AEs, SAEs, AEs that cause discontinuation from the study treatment, and AESIs (as described in Section 5) will be analyzed in a similar way to AEs in Phase–II. The summaries will include all patients who received at least one dose of study medication.

#### Randomized Phase II: Exploration of EfficacySafety: in mBC

#### Safety endpoints will be summarized by treatment group.

Safety endpoints during the Randomized Phase II part of the study will be assessed via: total AEs, AEs Grade ≥ 3, SAEs, premature withdrawal from study and study medication, AESIs, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

The incidence of AEs and SAEs will be summarized according to the primary system organclass (SOC) and within each SOC, by MedDRA preferred term. Time to onset of the first episode of AESI will also be summarized via Kaplan-Meier method. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry, will be presented in shift tables of NCI-CTC grade at baseline *versus* worst grade during treatment for the Randomized Phase II of the study, Cohort 1 and overall.

#### Phase-I, Cohort 2: MTD Finding: mGC

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

Safety parameters will be summarized in a similar way to Phase-I, Cohort 1: mBC.

#### **Exploratory Analyses**

For all patients a retrospective central confirmation of the HER2 status will be done. Further exploratory analysis for HER2-positive patients (based on central confirmation) will be done for selected endpoints, e.g. BOR and safety (AEs, SAEs, AEs with Grade ≥ 3, and AESIs).

Subgroup analysis for BOR, safety (AEs, SAEs-and AE, AEs with Grade ≥ 3, and AESIs) in the Randomized Phase–II part of the study will be presented for both treatment groups: elderly *versus* younger patients, patients with ECOG 0–1 *versus* ECOG 2. More details will be presented in the statistical analysis planSAP.

#### **Determination of Sample Size**

#### Sample Size for Phase-I: MTD Finding: mBC

This part will be based on a classical 3 byplus 3 Phase—I design. From 3A minimum of 6 and up to 18—patients mightwill be enrolled in Cohort—1. There is no formal sample size estimation for this part.

Sample Size for Randomized Phase—II: Exploration of Efficacy:—and Safety in mBC

Assuming a preferable BORR of 75% to 80% in Cohort 1 (mBC patients) and aiming for aprecision of 8 10%, lower limit of 95% confidence interval of at least 65%, a total of 100patients would need to be evaluable for Cohort 1.

Approximately 117 patients (78 patients in the combination of T-DM1 and capecitabine respective 39 patients in T-DM1 treatment group), including a 10% withdrawal rate, will be randomized with a 2:1 ratio to the combination of T-DM1 and capecitabine or T-DM1.

Point estimates and 95% Clopper-Pearson exact CIs are tabulated for a range of possible BOR outcomes for both treatment groups:

## Table 1: Sample Size Estimation (2:1 randomization)

| Total number of patient | <del>s is 100 (Phase II)</del> | |
|---|---|---|
| Number of Patients/ | 95% Clopper Pearson Confider | nce Intervals |
| Response | | |
| 75 patients (75%) | <del>65% 83 %</del> | |
| 80 patients (80%) | | <del>71% 87%</del> |
| Total number of patien | ts adjusted for 10% withdrawal ra | ate is 110 patients |

| N (T-DM1 and capecitabine)* = 70 patients* | |
|---|---|
| BOR rate [%] | 95% CI (within treatment group) [%] |
| <mark>57.5</mark> | <del>(45.1–69.2)</del> |
| <mark>60.0</mark> | <del>(47.6–71.5)</del> |
| <mark>62.5</mark> | (50.1–73.8) |
| <mark>65.0</mark> | (52.7–76.0) |
| <mark>67.5</mark> | (55.2–78.2) |
| N (T-DM1) = 35 patient | s* |
| BOR rate [%] | 95% CI (within treatment group) [%] |
| BOR rate [%]<br>37.0 | 95% CI (within treatment group) [%] (21.4–54.9) |
| 37.0 | |
| | (21.4–54.9) |
| 37.0<br>40.0 | (21.4–54.9)<br>(23.9–57.9) |
| 37.0<br>40.0<br>43.0 | (21.4–54.9)<br>(23.9–57.9)<br>(26.4–60.8) |

-BOR of 75% could be estimated to be within 65% and 83% with a probability of 95% (Clopper Pearson exact confidence intervals). Adjusting for a withdrawal rate of approximately 10%, 110 patients will be enrolled in this phase.

The BOR rate of 75% is chosen based on the previously published data with trastuzumaband capecitabine (see protocol for reference)

The estimation of Sample Size is performed by Nquery and SAS programs.

Expected BOR rate for patients who received trastuzumab emtansine of 43.6% (95% CI: 38.6% – 48.6%) was chosen based on previously published data for trastuzumab emtansine (see Section 6.1 of the main body of the protocol for reference).

The precision for the BOR estimate of the combination of T-DM1 and capecitabine is approximately 12%, e.g. BOR of 60%, 95% CI of (47.6%, 71.5%). Due to the lower sample size of the treatment group T-DM1, the corresponding precision for the BOR estimate is increased to 18%, e.g. BOR of 46%, 95% CI of (29.1%, 63.6%)

A 2:1 randomization will be applied to allow more patients being exposed to the combination of T-DM1 and capecitabine. This will enable a more thorough assessment of the corresponding safety profile.

#### Stratification Factors

The following stratification factor will be implemented in the Randomized Phase II part of the study:

Number of prior lines of treatment for metastatic disease (1 or >1; excluding single-agent hormones).

A treatment line is defined as any treatment regime given to patient from treatment initiation until confirmed disease progression.

Sample Size for Phase I, Cohort 2: MTD Finding: mGC

This part will be based on a classical 3 byplus 3 Phase—I design. From 3 to 4812 patients might be enrolled in Cohort—2.

# 1. BACKGROUND

## 1.2 BACKGROUND ON STUDY DRUGS

## 1.2.1 TRASTUZUMAB EMTANSINE

## 1.2.1.6 Phase—III Study TDM4370g

This study of trastuzumab emtansine, met both primary efficacy endpoints of PFS by independent review and OS in patients with mBC previously treated with a taxane and trastuzumab (HERCEPTIN).

This trial has met its co-primary endpoint of improving PFS (by independent review committee) compared to those who received the combination of lapatinib and capecitabine.

PFS was 9.6 months Patients in the trastuzumab emtansine arm had a median PFS of 9.6 months versus 6.4 months for patients in the control arm of lapatinib and + capecitabine arm. OS has not yet been reached (HR = 0.65; 95% CI: 0.55–0.77; p < 0.001, log-rank test). Patients in the trastuzumab emtansine arm while had a median OS of 30.9 months versus 25.1 months for patients in the control arm the OS was 23.3 months. The of lapatinib + capecitabine (HR for PFS was = 0.650 (68; 95% CI: 0.55, -0.7785; p =< 0.0001001, log-rank test).

It iswas concluded that overall, there is no concern regarding the clinical safety of trastuzumab emtansine for the patient population that was studied, based on the currently available data. (Verma et al. 2012).

# 1.3 STUDY RATIONALE AND RISK-BENEFIT RISK ASSESSMENT

# 1.3.1 FOR MBC

The Phase–III, TDM4370g trial met its co-primary endpoint of improving PFS (by IRC)IRB) and OS compared towith those who received the combination of lapatinib and capecitabine (see Section 0).1.2.1.6).

Approximately 20002,000 patients with breast cancer BC have been treated in trastuzumab emtansine clinical trials with an acceptable safety profile and a positive risk-benefit ratio. A safety monitoring is in place to avoid potential everlapping toxicities. A broad development program is in place to seek approval for indications for mBC. Capecitabine in combination with anti-HER2

agent is a proven efficacious regimen with a well-established safety profile in mBC. Trastuzumab emtansine and capecitabine have no known significant overlapping toxicities. As a part of the Phase I conduct, regular teleconference calls with the investigators will be held to discuss the study treatment risk-benefit profile for each patient. An IDMC will be established with the main responsibility to assess the risk-benefit for the Phase II part of the study.

## 1.3.2 FOR MGC

A development program for trastuzumab emtansine is in place to seek approval for mGC indications. Capecitabine in combination with anti-HER2 agent is a proven efficacious regimen with a well—established safety profile in mGC. Trastuzumab emtansine and capecitabine might have overlapping toxicities and therefore a safety monitoring is in place to avoid exposing patients to harm. Therefore, exploring the benefit of combination therapy of trastzumab emtansine and capecitabine in mGC patients with mGC seems justified. Results from the Phase I part of the study in mGC will be used as supporting information for future studies in the indication.

# 2. OBJECTIVES

# 2.2 RANDOMIZED PHASE II: EXPLORATION OF EFFICACY AND SAFETY IN MBC PATIENTS

### 2.2.1 PRIMARY OBJECTIVE

To explore the efficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine in patients with mBC, as measured by ORR by RECIST v.1.1 per investigator local assessment

## 2.2.2 SECONDARY OBJECTIVES

Safety profile of the combination atof trastuzumab emtansine and capecitabine compared with trastuzumab emtansine

To explore the dose established during Phase lefficacy of the combination of trastuzumab emtansine and capecitabine compared with trastuzumab emtansine in patients with mBC, as measured by:

- Time to response (TTR)
- Duration of response (DoR)
- Time to progression (DoR)
- TTP)
- Time to treatment failure (TTF)
- Progression free survival (PFS)
- Clinical benefit rate (CBR)
- Overall survival (OS)
- PFS
- CBR

## OS

# 3. <u>STUDY DESIGN</u>

### 3.1 DESCRIPTION OF STUDY

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine in a Phase–I study in bothpatients with mBC and locally advanced or mGC-patients. The MTD efficacy and safety of the combination in patients with mBC will also be assessed for anti-tumor effects-(exploration of efficacy)explored in a randomized, open-label Phase–II, single-arm part of the study in the mBC cohort. There will be no exploration of efficacy in the mGC cohort.

### 3.1.1 OVERVIEW OF STUDY DESIGN

## **Overview of Study Design**

The study is designed to determine the MTD of capecitabine in combination with trastuzumab emtansine, in patients with HER2-positive mBC and locally advanced or mGC patients, using a Phase—I design, followed by a randomized, open-label Phase—II single armpart of the study to explore the efficacy and safety of the combination in mBC patients with mBC. There will be no exploration of efficacy in the mGC cohort. Results from the Phase—I in mGC will be used as supporting information for future studies in the indication.

## **Duration of Treatment and Patient Follow-up**

<u>Length of treatment:</u> All patients will be treated until disease progression, intolerable toxicity, withdrawal of consent, or death.

<u>Patient follow-up:</u> All patients from both cohorts will be followed—up until intolerable toxicity, withdrawn consent, death, or up to a maximum of 2 years after the last patient was <u>enrolledrandomized</u> in the <u>Randomized</u> Phase—II part of the study, whichever occurs first.

# <u>Duration of Study, Data Base Database</u> Closure and Data Reporting

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to be 2 years for dose finding the Dose Finding and the Phase—II/-Exploration of Efficacy and Safety. The study will end after the follow-up period wasis completed, as defined above. Last patient last visit (LPLV) is defined as the last data collection point that can be either a clinic visit or a lablaboratory sample. At that time point, the database will be closed.

In the case that in Cohort—1 the dose level 1 Dose Level -2 is too toxic (> 1/3-or >1/6 of dose-limiting toxicity [DLT]), the combination may be considered unfeasible. Enrollment, recruitment will be closed and no other neither the Randomized Phase II nor mGC cohort will be opened. Patients, who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the Steering Committee (SC).

Data may be reported at the end of each cohort i.e., once the MTD for Cohort—1 for mBC has been defined and the dose for Phase—II/Exploration of Efficacy and Safety has been selected. The latest point to write the Clinical Study Report (CSR) will be one—1 year after database closure.

Figure 4 Overview of Study Design



<sup>&</sup>lt;sup>1</sup> Capecitabine doses are administered daily on daysDays 1 to 14 of the 3-week cycles

#### 3.1.1.1 Overview of Phase I Design in Patients with mBC

<sup>&</sup>lt;sup>2</sup> The MTD defined in mBC Phase–I will be implemented in mBC Randomized Phase–II and mGC Phase–I

<sup>&</sup>lt;sup>3</sup> Cohort–<sup>2</sup> will open to recruit mGC patients with mGC once the MTD is defined in Phase–I for mBC patients

<sup>&</sup>lt;sup>4</sup>Patients on MTD in Phase I must re-consent, recruitment with mBC. Dose Level 1 will not be extended to 110 mBC patients explored in Cohort 2 (see also Section 3.3.2.1)

mBC = metastatic breast cancer; mGC = metastatic gastric cancer; MTD = maximum tolerated dose; q3w = every 3 weeks; qw = weekly; T-DM1 = trastuzumab emtansine



Figure 5 Overview of Phase—I Dose Finding Study Design

<sup>1</sup>If Dose level 1 is too toxic (>1/3 or >1/6 DLT), the study will be terminated. DLT = dose limiting toxicity; MTD = maximum tolerated dose



<sup>&</sup>lt;sup>1</sup> Repeat with the new dose level until the MTD is established

DLT = dose-limiting toxicity; MTD = maximum tolerated dose

<sup>&</sup>lt;sup>2</sup> If Dose Level -2 is too toxic (> 1/6 DLT), the study will be terminated.

# Determination of the Maximum Tolerated Dose in mBC Patients with mBC

The trial will first investigate the feasibility of the combination of capecitabine and trastuzumab emtansine q3w in one cohort up to 18 patients, by deescalating the dose of capecitabine from 750 mg/m² bid to 1000-650 mg/m² bid on daysDays 1 to 14 in cycles of 3 weeks with a 3 byplus 3 classical Phase—I design. Cohort—I will open first and enroll patients with HER2-positive mBC.

#### **Enrollment into Cohort 1**

Dose finding in patients with mBC (Phase I)

If dose level 1Dose Level -2 is found to be too toxic (DLT >1/3 or > 1/6), the enrollment combination may be considered unfeasible, the recruitment will be closed and the study will be terminated. neither the Randomized Phase II nor mGC cohort will be opened. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the SC.

The following escalation MTD determining rules will be applied during the dose finding Dose Finding treatment phase:

- Step 1: Three patients will be enrolled at dose level Dose Level 1
- Step 2: The toxicity of dose level Dose Level 1 will be monitored and the following actions taken:
  - a) If none of these three 3 patients (0/3) experiences a DLT, escalation to dose level 2 will occur the MTD will be established as the current dose level and will need to be confirmed in 3 more patients (to achieve ≤ 1/6 DLT at the current dose level)
  - b) If one1 of the initial three3 patients (1/3) experiences a DLT, an additional three3 patients should be enrolled and treated at the same dose, i.e. dose level., Dose Level 1
  - c) If no more patients experience a DLT (1/6), escalation to the nextMTD will be established as the current dose level will occur
  - d) If ene1 or more patients experience a DLT (> 1/6), the MTDdose will be established asde-escalated to the immediate inferiornext lower dose level or the study may be terminated if it happens at dose level 1. If no more than 1 patient experiences a DLT (≤ 1/6) after dose de-escalation, the dose will be considered the MTD and, following iDMC agreement, will be further explored in the Randomized Phase II part of the study. Dose re-escalation will not be allowed. If 2 or more patients experience DLT (> 1/6) after dose de-escalation, de-escalation should continue to the next lower dose level. Based on the DLT findings, the next dose level may be considered the MTD and, following iDMC agreement, be further explored in the Randomized Phase II part of the study or the study may be terminated if > 1/6 DLTs occur at Dose Level -2

- Step 3: Step 2 should be repeated until the MTD is reached
- If the last dose exceeds the MTD, de escalation to the previous dose should occur. This dose should be defined as MTD if 6 or more patients have been safely treated at this dose level and no more than 1/6 of the patients experienced a DLT at that dose level.
- If only 3 patients have been treated at this dose level, then 3 more patients will be treated and observed at this level in order to achieve at least 6 patients treated at the same dose level.

In order to define the dose for the Randomized Phase II/exploration Exploration of efficacy Efficacy and Safety part of the study, the Steering Committee will evaluate not only the DLTs during Cycle 1 will be evaluated but also all available safety information during the subsequent cycles. The dose level considered optimal by the Steering Committee will be the dose level selected to move forward with in the Phase II and mGC parts of the study.

Once the appropriate dose of study medication is established, the other cehorts Randomized Phase II part of the study and Phase I, Cohort 2 will open as per Figure 4.

# 3.1.1.2 Overview of Phase II: Exploration of Efficacy and Safety in Patients with mBC

This part of the study will explore the efficacy and safety of the combination treatment of T-DM1 and capecitabine, at the established MTD, compared with T-DM1 alone in mBC patients.

Once the Steering Committee MTD has been defined the MTD to treat patients in Phase II, approximately 117 additional 90 100 mBC patients will be enrolled.

Only the mBC patients who have received the MTD dose from Phase I with mBC will continue with be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to assess efficacy and safety of this treatment combination of capecitabine and trastuzumab emtansine. the Phase II part of the study; however, they will be followed-up until end of study (EOS).

Patients will be treated until disease progression/recurrence, intolerable toxicity, withdrawn consent, or death. If capecitabine needs to be discontinued for any reason, trastuzumab emtansine may continue, and the patient will be followed-up until EOS. In case of discontinuation of trastuzumab emtansine, patients will be followed-up until EOS.

All patients will be followed-up until withdrawn consent, death, or up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first.

See Section 3.1.1 for further information.

# 3.1.1.3 Overview of Phase I Design in mGC Patients

#### **Enrollment into Cohort 2**

The dose levels for escalation or de-escalation of capecitabine will be the same as described for Cohort—1; except for Dose Level 1, which will not be explored in patients with mGC (see also Section 3.3.2.1).

If the MTD established in Cohort–1 wasis defined at Dose Level -1:

- This will be the starting dose level 1 of 750 mg/m² bidin Cohort 2. If Dose Level -1 is well tolerated (DLT ≤ 1/6), this dose will be established as the MTD for mGC.
  - If dose level 1 is tolerated, doses should be escalated to dose level 2 of 850 mg/m²-bid
- If dose level De-escalation: if Dose Level -1 is not tolerated (>1/3-or>in Cohort 2 (> 1/6 DLT), de-escalation will be to Dose Level -2.

If the MTD established in Cohort 1 is defined at Dose Level -2:

- This will be the starting dose in Cohort 2. If Dose Level -2 is well tolerated (DLT ≤ 1/6), this dose will be established as the MTD for mGC.
- De-escalation: if Dose Level -2 is not tolerated in Cohort 2 (> 1/6 DLT), the combination will be considered not feasible in mGC and Cohort— 2 will be terminated. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the SC
- e) If the MTD in Cohort 1 was defined at dose level 2 of 850 mg/m<sup>2</sup> bid
  - If dose level 2 is tolerated, doses should be escalated to dose level 3 of 1000 mg/m²-bid
  - If dose level 2 is not tolerated, doses should be de escalated to doselevel 1 of 750 mg/m²-bid
- f) If the MTD in Cohort 1 was defined at dose level 3 of 1000 mg/m<sup>2</sup> bid
  - If dose level 3 is tolerated, no escalation will be done and the MTDwill be defined at dose level 3

# 3.1.1.4 Considerations for all Patients Treated in the Study

Safety data will be reviewed on an ongoing basis (i.e. real time safety monitoring) by the Steering Committee. The preliminary safety review will be based on the safety information (DLTs, dose delays, dose reductions and Grade 3 5 events) observed during the first cycle in at least 3 patients.

#### 3.1.1.5 Number of Patients

Overall, it is anticipated that the maximum number of patients enrolled into the study will be 440approximately 147 patients.


## Phase-I, Cohort 1: mBC

From 3—a minimum of 6 to 18 patients will be enrolled into Cohort—1 to determine the MTD of capecitabine in combination with trastuzumab emtansine in mBC—patients with mBC.

## Randomized Phase-II: Exploration of Efficacy and Safety in mBC

For this part of the study, Cohort 1 a total of approximately 117 patients with mBC will be expanded to 110 mBC patients randomized.

## Phase-I, Cohort 2: mGC

After the MTD in Cohort—1 has been established, 3—1812 patients will be enrolled into Cohort—2 to determine the MTD of capecitabine in combination with trastuzumab emtansine in mGC patients with mGC.

# 3.1.2 STEERING COMMITTEE

A Steering Committee A SC has been established for this study. Initially, it is composed of the investigators participating in the Phase-I, Cohort-1 part of the study and one medical representative and one statistician of the Sponsor. The study design and DLT has been developed by the Steering Committee.

See Steering Committee SC. See SC Charter for further information.

The SC will collectively review the status of the ongoing patients on a regular basis. The SC will also review in due course all available efficacy data and PK information to ensure that safety information is in the context of risk-benefit and that dosing is also related to exposure to the drug.

The SC will adjudicate in cases of DLTs that are not covered by the existing DLT criteria.

## 3.1.3 INDEPENDENT DATA MONITORING COMMITTEE

An independent data monitoring committee (IDMC) will be established for the Randomized Phase II part of the study. The IDMC will review the safety outcomes for patients enrolled in Phase I, Cohort 1 and advise whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 20 and 60 patients have received at least 3 cycles (Cycle 3 Day 1) of treatment in the Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II of the study or as requested.

#### 3.2 END OF STUDY

End of study (EOS) is defined as LPLV at the end of the follow-up period, as defined in Section 3.1.1. This will be the last data collection point, which can be a clinic visit or a laboratory sample. LPLV is expected to occur approximately 2 years after the last patient has been enrolled into the trial.

## 3.3 RATIONALE FOR STUDY DESIGN

# 3.3.1 RATIONALE FOR PATIENT GROUP SELECTION

#### 3.3.1.1 Rationale for Phase I

Following review of preliminary data from Cohort 1 of this study by the SC for patients enrolled to receive 750 mg/m<sup>2</sup> capecitabine, where 2 DLTs were observed in 6 evaluable patients, it was decided not to explore dose levels of capecitabine higher than 750 mg/m<sup>2</sup>. According to the investigator assessment and the SC recommendation, the available evidence shows an acceptable positive risk-benefit in all 7 patients treated at Dose Level 1.

As of 7 August 2013, five patients remain on treatment, with a follow-up period of 4 to 8 months. Of the two patients who have discontinued treatment, one patient's disease has progressed, and the other discontinuation was based on the investigator's decision, following the central confirmation, that the patient's disease was HER2-negative. Considering the available safety data for all patients (maximum number of cycles is 12), the combination of capecitabine and T-DM1 is well tolerated, except for increases in transaminases and hand-foot syndrome. Dose modifications of T-DM1 and/or capecitabine have allowed those patients to continue on treatment. Of note, no SAE has been reported in 6 patients. Latest tumor response data show 2 patients with PR and 4 patients with SD. Any required dose modifications (dose reductions) are allowed for each individual drug as described in Sections 5.1.5.1 and 5.1.5.2 and are in line with the trastuzumab emtansine Investigator's Brochure and Xeloda® Summary of Product Characteristics.

The combination of T-DM1 and capecitabine will be evaluated with a deescalation study design. Patients who are currently receiving the combination of T-DM1 and capecitabine 750 mg/m<sup>2</sup> can continue to receive the dose as per protocol until there is no longer evidence of positive risk-benefit as per investigator assessment and SC endorsement.

#### 3.3.1.2 Rationale for Randomized Phase II

Randomized Phase—II II part of the study is designed to provide an estimation of the treatment effect of the combination, at the selected MTD—, compared with T-DM1 alone.

The patient data will be stratified by previous anti-cancer treatment (excluding single-agent hormones) for the treatment of metastatic disease (1 or >1prior lines of treatment). The stratified data will be compared with data from historical studies of single-agent trastuzumab emtansine in similar patient populations. This will allow a more robust evaluation of the added treatment effect of Xeloda® within the combination treatment.

A 2:1 randomization will be applied to allow more patients being exposed to the combination of T-DM1 and capecitabine. This will enable a more thorough assessment of the corresponding safety profile.

# 3.3.2 RATIONALE FOR INVESTIGATIONAL MEDICINAL DOSE SELECTION

#### 3.3.2.1 In Patients with mBC

Capecitabine doses have been selected as being in the range of efficacious doses for single—agent or combination use. The dosedoses selected are within the dosing range included in the Xeloda® Summary of 750 mg/m²-bidwasProduct Characteristics (SmPC) and therefore are considered the minimum to be efficacious dose. The maximum dose of 1000 mg/m²-bid is the currently approved dose of capecitabine (please see the current national prescribing information of Xeloda®)..

#### 3.4 OUTCOME MEASURES

## 3.4.1 PHASE—I: MBC

## 3.4.1.3 Primary Safety Outcome Measure

The primary safety outcome measure is to establish the MTD. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination and will be summarized for each treatment dosage.

# 3.4.1.4 Secondary Safety Outcome Measures

Safety endpoints will be summarized for both treatment phases: dose findingand exploration of efficacy. Again, the summary of safety endpoints will be presented for each cohorteach treatment dosage:

- Incidence, nature and severity of AEs, as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v. 4.0
- Incidence, nature, and severity of serious SAEs, as per NCI CTCAE v. 4.0
- Incidence and nature of AEs equal or higher than Grade 3
- Incidence, nature, and severity of AEs of special interest (AESIs), as per NCI CTCAE v. 4.0
- Premature withdrawal from study and study medication
- Abnormal laboratory values
- LVEF
- Exposure to study medication
- Concomitant medications and physical examination

# 3.4.2 RANDOMIZED PHASE II: EXPLORATION OF EFFICACY AND SAFETY IN MBC

## 3.4.2.1 Primary Efficacy Outcome Measure

The primary outcome measure is ORR by investigator assessment, based on best overall response (BOR) (defined as the best response recorded from the start of treatment randomization into Phase II part of the study and until

disease progression or frecurrence, or death, withdrawal of consent, or EOS, whichever occurs first; or for newly enrolled patients the best response from the start of Phase II until disease progression or death) by investigator assessment; as per RECIST v.1.1 provided in Appendix 3.

## 3.4.2.3 Primary Safety Outcome Measure

A primary safety outcome is defined only for Phase I, and will be presented for both treatment groups.

## 3.4.2.4 Secondary Safety Outcome Measures

Safety endpoints will be summarized for both treatment phases: dose finding and exploration of efficacy. Again, the summary of safety endpoints will be presented for each cohort:

- Incidence, nature and severity of AEs, as per NCI CTCAE v. 4.0
- Incidence, nature, and severity of serious SAEs, as per NCI CTCAE v. 4.0
- Incidence and nature of AEs equal or higher than Grade 3
- Incidence, nature, and severity of AESIs, as per NCI CTCAE v. 4.0
- Premature withdrawal from study and study medication
- Abnormal laboratory values
- LVEF
- Exposure to study medication
- Concomitant medications and physical examination

## 3.4.3. PHASE I: MGC

## 3.4.3.3 Primary Safety Outcome Measure

The primary outcome measure is to establish MTD. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination and will be summarized for each treatment dosage.

#### 3.4.3.4 Secondary Safety Outcome Measures

Safety endpoints will be summarized for both treatment phases: dose finding and exploration of efficacy. Again, the summary of safety endpoints will be presented for each cohort:

- Incidence, nature and severity of AEs, as per NCI CTCAE v. 4.0
- Incidence, nature, and severity of serious SAEs, as per NCI CTCAE v. 4.0
- Incidence and nature of AEs equal or higher than Grade 3.
- Incidence, nature, and severity of AESIs, as per NCI CTCAE v. 4.0
- Premature withdrawal from study and study medication
- Fatal cases and causes of death
- Abnormal IL aboratory values

- LVEF
- Treatment Eexposure to study medication
- Concomitant medications and physical examination

# 4. MATERIALS AND METHODS

#### 4.1 PATIENTS

#### 4.1.3 INCLUSION CRITERIA

### 4.1.3.1 For mBC Patients with mBC

- 8. Liver function:
  - a) Total bilirubin ≤ 1.5 × upper limin of normal (ULN) except in patients with previously documented Gilbert's syndrome in which case total bilirubin ≤ 3 mg/dL is acceptable
  - d) Evidence of stable liver function during the month prior to enrollment with liver function tests' (LFTs) fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN

#### 4.1.3.2 For Patients with mGC

- 8. Liver function:
  - a) Total bilirubin ≤ 1.5 × ULN except in patients with previously documented Gilbert's syndrome in which case total bilirubin ≤ 3 mg/dL is acceptable
  - d) Evidence of stable liver function in the month prior to enrollment with LFTs fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN
- 11. Histologically or cytologically confirmed mGC or locally advanced GC

# 4.1.4 EXCLUSION CRITERIA

#### 4.1.4.1 For mBC Patients: with mBC

- 6. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product
- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 360-500 mg/m<sup>2</sup>
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 360-500 mg/m² doxorubicin.

23. No signs and symptoms suggestive that the patient has dihydropyrimidine dehydrogenase (DPD) deficiency

#### 4.1.4.2 For Patients with mGC

- 7. History of exposure to the following cumulative doses of anthracyclines:
  - a) Doxorubicin or liposomal doxorubicin > 360-500 mg/m²
  - d) If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 360-500 mg/m<sup>2</sup> doxorubicin.
- 22. No signs and symptoms suggestive that the patient has DPD deficiency
- 23. Lapatinib ≤ 14 days before first study drug administration

# 4.1.5 PATIENT REPLACEMENT POLICY

None of the patients in the Phase I part of the study may be replaced unless approved by the entire SC.

### 4.2 METHOD OF TREATMENT ASSIGNMENT

In the Randomized Phase II part of the study, patients will be randomized to receive either the combination of T-DM1 and capecitabine or T-DM1 alone. The 2:1 randomization ratio will be applied to allow more patients being exposed to the combination treatment and to enable a more thorough assessment of the corresponding safety profile.

This is an open-label study; therefore, no blinding will be used.

## 4.3 STUDY TREATMENT

#### 4.3.2 DOSAGE AND ADMINISTRATION

## 4.3.2.1 For Patients with mBC

#### **Trastuzumab Emtansine**

The first infusion of trastuzumab emtansine will be administered over 90 minutes (±10 minutes). Infusions may be slowed or interrupted for patients experiencing infusion—associated symptoms. Vital signs must be assessed before and after dose administration. Following the initial dose, patients will be observed for at least 6090 minutes for fever, chills, or other infusion—associated symptoms.

### Capecitabine

Capecitabine will be administered twice a day, orally for 14 days followed by a 7-day rest period at the dose levels Dose Levels 1—3 to -2 described in the "study design" Section ..3.1.1. Capecitabine tablets should be swallowed with water within 30

minutes after a meal. Capecitabine doses can be delayed for up to 4 hours, while keeping the minimal interval of 8 hours between the doses.

Rounding of the dose, based on 150 and 500 mg strength tablets, will be allowed to the nearest dose per patient body surface area (BSA).

If a dose is missed, the patient should skip that dose. The patient should not double the dose during the next administration.

For Phase II, guidelines Guidelines for dosage modification and treatment interruption or discontinuation are provided in Section ..5.1. For this part of the study, the MTD fromestablished in Phase-II, Cohort 1 will be used as a starting dose.

### 4.3.2 2 For mGC Patients with mGC

### Capecitabine

Capecitabine will be administered twice a day, orally, for 14 days followed by a 7-day rest period at the dose level that was determined during the dose finding Dose Finding part of the study in mBC patients with mBC as the MTD in Cohort—1. Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Capecitabine doses can be delayed for up to 4 hours, while keeping the minimal interval of 8 hours between the doses.

#### 4.5 STUDY ASSESSMENTS

## 4.5.1 DESCRIPTION OF STUDY ASSESSMENTS

## 4.5.1.4 Tumor and Response Evaluations

Measurable and unmeasurable disease must be documented at screening and re-assessed at each subsequent tumor evaluation. Tumor assessments with computed tomography (CT) or magnetic resonance imaging (MRI) scans of the chest, abdomen, and pelvis are to be performed as described in Appendix 1, Schedule of Assessment. CT or MRI of the brain and baseline radioisotope bone scan must be obtained at screening. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to first treatment the bone scan does not need to be repeated and non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Tumor assessments should include an evaluation of all known and/or suspected sites of disease, whenever possible. Patients should have lesions selected that can be evaluated at every tumor assessment. The same radiographic procedure used at screening must be used throughout the study (e.g., the same contrast protocol for CT scans). Response assessments will be assessed by the investigator, based on physical examinations, CT or MRI scans, and bone scans using RECIST v. 1.1 (see ). In the event a positron emission tomography (PET)/CT scanner is used for tumor assessments, the CT portion of the PET/CT must meet criteria for diagnostic quality. Please consult the Imaging Manual for guidelines on performing a diagnostic quality (optimized) CT exam. For patients who continue study treatment after isolated brain progression, the frequency of follow-up scans is at the discretion of the investigator.

### 4.5.1.5 Laboratory Assessments

## **Local Laboratory Assessments:**

- Hematology, biochemistry, coagulation, urinalysis, and pregnancy testing
- Prospective or retrospective HER2 status. Patients will be enrolled based on local results.

### **Central Laboratory Assessments:**

 Retrospective HER2 status. Retrospective central confirmation will not impact the treatment decisions or primary endpoint of Phase I, Cohort 1 and will be used to validate efficacy analyses in Phase I and to censor the efficacy population for the Randomized Phase II part of the study

#### 4.5.1.7 ECOG Performance Status

Performance status will be measured using the ECOG performance status scale (see Appendix 6).

It is recommended, where possible, that a patient's performance status be assessed by the same person throughout the study.

Performance status will be assessed according to the schedule of assessments (see Appendix 1)

### 4.5.2 TIMING OF STUDY ASSESSMENTS

#### 4.5.2.1 Screening and Pretreatment Assessments

Results of standard of care tests or examinations performed prior to obtaining informed consent and within 28 days prior to study start may be used; such tests do not need to be repeated for screening. Patient must have stable liver tests prior to the first dose of study drug.

Patients who are on the MTD dose established in Cohort 1 will not contribute to Phase II; however, they will be followed-up until end of studyEOS. In Randomized Phase II, patients will be randomized in a 2:1 ratio to receive T-DM1 or the combination of T-DM1 and capecitabine prior to receiving the first dose of study medication.

Patients who are on the MTD dose established in Cohort 1 must re consent to be enrolled into Phase II.

Patients in Cohort 1 will not contribute to Phase II; however, they will be followed-up until EOS. In Randomized Phase II, patients will be randomized in a 2:1 ratio to receive

T-DM1 or the combination of T-DM1 and capecitabine prior to receiving the first dose of study medication.

## 4.5.2.3 Assessments at Study Completion/Early Termination Visit

Patients may remain on study treatment until disease progression as assessed by the investigator, intolerable toxicity, or until the patient wishes to withdraw from study treatment. Patients who discontinue study treatment will

be followed-up until EOS and will be asked to return to the clinic approximately 28–42 days after the last study treatment administration, for the safety follow-up visit.

# 4.6 PATIENT, STUDY, AND SITE DISCONTINUATION

#### 4.6.1 PATIENT DISCONTINUATION

Patients must be withdrawn from study treatment if they become pregnant or experience any of the following:

### Pregnancy

Disease disease progression defined using RECIST v. 1.1 Appendix 3. The exception to this is patients who develop isolated progression in the brain as described in Appendix 3.

Unacceptable Details of discontinuation due to toxicity because of the trastuzumab emtansine dose as specified are given in Section 5.1.

 Unacceptable toxicity because of the capecitabine dose as specified in Section 

Other reasons for patient discontinuation may include, but are not limited to, the following:

- Noncompliance
- Pregnancy
- Non-compliance
- Investigator decision based on the patient's best interest
- Patient decision

# 5. ASSESSMENT OF SAFETY

## 5.1 SAFETY PLAN

All patients will be monitored closely for toxicity. The potential important safety issues anticipated in this trial, as well as measures intended to avoid or minimize such toxicities, are outlined in the following sections.

#### 5.1.1 RISKS ASSOCIATED WITH TRASTUZUMAB EMTANSINE

Trastuzumab emtansine dose modifications are described in Section .

The following summarizes the experience with trastuzumab emtansine inmultiple breast cancer studies to date. Trastuzumab emtansine has demonstrated a favorable toxicity and tolerability profile to date acrossmultiple studies. Please refer to the Investigator's Brochure for furtherinformation.


Reversible thrombocytopenia has been commonly observed in completed and ongoing studies with trastuzumab emtansine. Most events were Grade 1–2; Grade 3–4 thrombocytopenia has been observed less commonly. The incidence of Grade 1 thrombocytopenia gradually increased over successive cycles; however, there was no increase in the proportion of Grade ≥ 3-abnormalities. The number of patients who experienced platelet count recovery to normal levels by Day 1 of the subsequent cycle decreased with successive cycles, suggesting a modest cumulative effect of trastuzumab emtansine on platelet count. There was no clear association between thrombocytopenia and severe hemorrhagic events; however, the use of platelet transfusions has been reported.

Transient and reversible increases in serum AST and ALT have been observed across the trastuzumab emtansine studies. Grade 1–2 events have been observed frequently; Grade 3–4 events have been observed much less-commonly. The incidence of increased AST was substantially higher than that for ALT. Increases in AST and ALT were commonly observed by Day 8 of each cycle and generally returned to baseline by Day 21. The proportion of patients with Grade 1–2 increases in transaminases increased with-successive cycles; however, no increase in the proportion of Grade 3-abnormalities over time was observed. To date, there have been no cases meeting Hy's Law criteria for drug induced liver injury. Although significant hepatotoxicity has rarely been seen in clinical trials with trastuzumab-emtansine to date, the relationship to trastuzumab emtansine has not been established. Nevertheless, severe liver injury remains an important potential risk.

Infusion related reactions are known to occur with the administration of monoclonal antibodies and have been reported with trastuzumab emtansine. Infusion reaction AEs occurred rarely and were mostly Grade 1–2. Non-specific symptoms that occurred on the first day of trastuzumab emtansine infusion that could be associated with an infusion reaction included fatigue, nausea, chills, pyrexia, and, less commonly, headache, hypertension, vomiting, and cough.

Pneumonitis has been rarely reported with trastuzumab emtansine. Signs, symptoms, and clinical findings include dyspnea, cough, fatigue, and pulmonary infiltrates. There were no fatalities among the cases of pneumonitis reported with trastuzumab emtansine.

In clinical trials with trastuzumab emtansine, peripheral neuropathy has been reported, mainly as Grade 1 toxicity. Hypokalemia and decreases in serum potassium have been reported in completed and ongoing studies with trastuzumab emtansine. Most of these AEs were Grade 1–2.

Although significant cardiac events have been infrequent in clinical trials with trastuzumab emtansine to date, severe cardiotoxicity remains an important potential risk. Treatment with trastuzumab, a component of trastuzumab emtansine, has resulted in subclinical and clinical cardiac failure manifesting as CHF, decreased LVEF, and cardiac death. The incidence and severity of cardiac dysfunction was highest in patients who received trastuzumab concurrently with anthracycline containing chemotherapy regimens.

Cardiotoxicity, manifesting as a decline in LVEF or CHF, is being closely monitored in the trastuzumab development program. Across studies—TDM4258g, TDM4374g, and TDM4688g, approximately 273 patients were-treated, and a total of 8 patients recorded an asymptomatic decrease in baseline LVEF of at least 10%, concomitant with an LVEF < 50%. Two-patients had trastuzumab emtasine treatment withdrawn because of decreased LVEF. Rare cases of Grade 3 cardiac dysrhythmias have been reported among patients receiving trastuzumab emtansine, although a direct relationship to study drug remains unclear.

Importantly, preliminary evaluations of safety in the randomized study—TDM4450g suggest that the safety and tolerability of trastuzumab emtansine-compared favorably with that of trastuzumab plus docetaxel, with the overall-incidence of Grade ≥ 3 AEs favoring the trastuzumab emtansine arm (46.4%-vs. 89.4%) (data on file).

Full details regarding the clinical safety of trastuzumab emtansine are presented in Sections 5 and 6 of the Investigator's Brochure.

## 5.1.1.1 Cardiotoxicity

Patients treated with trastuzumab emtansine are at increased risk of developing left ventricular dysfunction. LVEF < 40% has been observed in patients treated with trastuzumab emtansine. Patients without significant cardiac history and with an LVEF ≥ 50% determined by ECHO or MUGA scan are eligible for study participation. LVEF will be monitored at screening and regularly throughout the study until the assessment at the safety follow-up visit. Patients with symptomatic cardiac dysfunction will be discontinued from study treatment. Asymptomatic LVEF declines will be handled as per the algorithm shown in Figure 6. Treatment with trastuzumab emtansine has not been studied in patients with LVEF < 50%.

#### 5.1.1.2 Hematologic Toxicity (Thrombocytopenia)

Thrombocytopenia, or decreased platelet counts, was reported in patients in clinical trials of trastuzumab emtansine. The majority of these patients had Grade 1 or 2 events (≥ 50,000/mm³), with the nadir occurring by Day 8 and generally improving to Grade 0 or 1 (≥ 75,000/mm³) by the next scheduled dose. In clinical trials, the incidence and severity of thrombocytopenia were higher in Asian patients. Severe cases of both non-fatal and fatal hemorrhagic events including central nervous system hemorrhage have been reported in clinical trials with trastuzumab emtansine; these events were independent of the patients' ethnicity. In some of the observed cases the patients were also receiving anti-coagulation therapy. The need for platelet transfusions has been reported.

Patients with thrombocytopenia and on anti-coagulant treatment have to be monitored closely during treatment with trastuzumab emtansine. Platelet counts will be monitored prior to each trastuzumab emtansine dose.

Use of erythropoiesis-stimulating agents will be allowed as consistent with prescribing guidelines. Transfusion of red blood cells and/or platelets will be allowed according to and at the discretion of the treating physician.

# 5.1.1.3 Hepatotoxicity

Hepatotoxicity, predominantly in the form of asymptomatic increases in the concentrations of serum transaminases (Grade 1 – 4 transaminitis), has been observed in patients while on treatment with trastuzumab emtansine in clinical trials. Transaminase elevations were generally transient. The incidence of increased AST was substantially higher than that for ALT. The proportion of patients with Grade 1 or 2 increases in transaminases increased with successive cycles, suggesting a modest cumulative effect of trastuzumab emtansine on transaminases; however, no increase over time in the proportion of Grade 3 abnormalities was observed. Patients with elevated transaminases improved to Grade 1 or normal within 30 days of the last dose of trastuzumab emtansine in the majority of the patients.

Rare cases of severe hepatotoxicity, including death due to drug-induced liver injury and associated hepatic encephalopathy, have been observed in patients treated with trastuzumab emtansine. While there is evidence of drug-induced liver toxicity (predominantly in the form of asymptomatic increases in the concentrations of serum transaminases) in patients treated with trastuzumab emtansine, its potential to cause acute severe liver injury with clinically meaningful changes in liver function is unclear as the observed cases of acute liver injury were confounded by concomitant medications with known hepatotoxic potential and/or underlying conditions. Nevertheless, a contributory role of trastuzumab emtansine in these cases cannot be excluded. Therefore, acute severe liver injury (Hy's law) remains an important potential risk with trastuzumab emtansine. A Hy's law case has the following components:

- Aminotransferase enzymes (ALT/AST) greater than 3 × ULN with concurrent elevation of serum total bilirubin to > 2 × ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)
- No other reason can be found to explain the combination of increased aminotransferases and serum total bilirubin, such as viral hepatitis A, B, or C, pre-existing or acute liver disease, or another drug capable of causing the observed injury
- The finding should be serious as shown by gross jaundice, clinical disability, need for hospital care, and be at least probably drug-induced (by trastuzumab emtansine)

Trastuzumab emtansine treatment in patients with serum transaminases  $> 3 \times \text{ULN}$  and concomitant total bilirubin  $> 2 \times \text{ULN}$  should be permanently discontinued.

Patients must have adequate and stable liver function: hepatic transaminases (AST/ALT) and total bilirubin must be within acceptable range, as defined in the protocol, within 4 weeks prior to the first dose of trastuzumab emtansine. Liver function will be monitored prior to each trastuzumab emtansine dose.

Cases of nodular regenerative hyperplasia (NRH) of the liver have been identified from liver biopsies in patients treated with trastuzumab emtansine and presenting with signs and symptoms of portal hypertension. NRH was also observed in one fatal case of hepatic failure. NRH is a rare liver condition characterized by widespread benign transformation of hepatic parenchyma into small regenerative nodules; NRH may lead to non-cirrhotic portal hypertension. Diagnosis of NRH can only be confirmed by histopathology.

NRH should be considered in patients who develop clinical symptoms of portal hypertension and/or a cirrhosis-like pattern seen on CT scan of the liver but with normal transaminases and no other manifestations of cirrhosis or liver failure following long-term treatment with trastuzumab emtansine. Upon diagnosis of NRH, trastuzumab emtansine treatment must be permanently discontinued.

# 5.1.1.4 Pulmonary Toxicity

Cases of interstitial lung disease (ILD), including pneumonitis, some leading to acute respiratory distress syndrome or fatal outcome, have been reported in clinical trials with trastuzumab emtansine. Signs and symptoms include dyspnea, cough, fatigue, and pulmonary infiltrates. These events may or may not occur as sequelae of infusion reactions. Treatment has included administration of steroids and oxygen, and study drug discontinuation. Patients with dyspnea at rest due to complications of advanced malignancy and comorbidities may be at increased risk of pulmonary events.

Treatment with trastuzumab emtansine has to be permanently discontinued in patients who are diagnosed with ILD or pneumonitis.

## 5.1.1.5 Infusion-related Reactions/Hypersensitivity

Infusion-related reactions characterized by one or more of the following symptoms, flushing, chills, pyrexia, dyspnea, hypotension, wheezing, bronchospasm, and tachycardia may occur with the administration of monoclonal antibodies and have been reported with trastuzumab emtansine. In general, these symptoms were not severe. In most patients, these reactions resolved over the course of several hours to a day after the infusion was terminated. Patients should be observed closely for infusion-related reactions, especially during the first infusion.

Patients should be observed closely for hypersensitivity. Serious, allergic/anaphylactic-like reactions have been observed in clinical trials with treatment of trastuzumab emtansine. Administration of trastuzumab emtansine will be performed in a setting with access to emergency facilities and staff who are trained to monitor and respond to medical emergencies. Patients will be observed closely for infusion-related/hypersensitivity during and after each trastuzumab emtansine infusion for a minimum of 90 minutes after the first infusion and for a minimum of 30 minutes after subsequent infusions in the absence of infusion-related AEs. Pre-medication is allowed according to standard practice guidelines. In the event of a true hypersensitivity reaction (in which severity of reaction increases with subsequent infusions), trastuzumab emtansine treatment must be

permanently discontinued. Patients who experience a Grade ≥ 3 allergic reaction or acute respiratory distress syndrome will be discontinued from study treatment.

### 5.1.1.6 Neurotoxicity

DM1, an anti-microtubule agent, can potentially cause peripheral neuropathy. Peripheral neuropathy, mainly Grade 1 and predominantly sensory, has been reported in clinical trials of trastuzumab emtansine. Treatment with trastuzumab emtansine should be temporarily discontinued in patients experiencing Grade 3 or 4 peripheral neuropathy until symptoms resolve or improve to  $\leq$  Grade 2. Patients should be examined for signs of peripheral neuropathy prior to each dose of trastuzumab emtansine. Patients who experience Grade  $\geq$  3 neurotoxicity in the form of peripheral neuropathy that does not resolve to Grade  $\leq$  2 within 42 days after last dose received will be discontinued from study treatment.

#### 5.1.1.7 Extravasation

In trastuzumab emtansine clinical studies, reactions secondary to extravasation have been observed. These reactions were usually mild and comprised erythema, tenderness, skin irritation, pain, or swelling at the infusion site. Rare reports of more severe events such as cellulitis, pain (tenderness and burning sensation), and skin irritation have been received as part of the continuing surveillance of trastuzumab emtansine safety. These reactions have been observed more frequently within 24 hours of infusion. Specific treatment for trastuzumab emtansine extravasation is unknown at this time. The infusion site should be closely monitored for possible subcutaneous infiltration during drug administration.

#### 5.1.1.8 Trastuzumab Emtansine Dose Modification

Trastuzumab emtansine dose modifications are described in Section 5.1.5.1.

## 5.1.2 RISKS ASSOCIATED WITH CAPECITABINE

Capecitabine dose modifications will be done according to Section , study design.

Patients treated with capecitabine should be carefully monitored for toxicity. Most AEs are reversible and do not require permanent discontinuation of therapy (please refer to the Xeloda<sup>®</sup> Investigator`s Brochure for more information).

The spectrum of cardiotoxicity observed with capecitabine is similar to that of other fluorinated pyrimidines. This includes myocardial infarction, angina, dysrhythmias, cardiac arrest, cardiac failure and electrocardiographic changes. These AEs may be more common in patients with a prior history of coronary artery disease.

DPD deficiency, a rarelyA rare, unexpected, severe toxicity (e.g. stomatitis, diarrhea, neutropenia, and neurotoxicity) associated with 5-FU has been attributed to a deficiency of dihydropyrimidine dehydrogenase (DPD)DPD

activity. Therefore, a link between decreased levels of DPD and increased, potentially fatal, toxic effects of 5-FU cannot be excluded.

Capecitabine can induce hand—foot syndrome (palmar-plantar erythrodysesthesia or chemotherapy-induced acral erythema), which is a cutaneous toxicity. For patients receiving capecitabine monotherapy in the metastatic setting, the median time to onset was 79 days (range 11-to—360 days), with a severity range of Grades 1 to 3. Grade 1 hand-foot syndrome is defined by numbness, dysesthesia/paresthesia, tingling or erythema of the hands and/or feet and/or discomfort which does not disrupt normal activities. Grade 2 is defined as painful erythema and swelling of the hands and/or feet and/or discomfort affecting the patient's activities of daily living (ADL). Grade 3 is defined as moist desquamation, ulceration, blistering or severe pain of the hands and/or feet and/or severe discomfort that causes the patient to be unable to work or perform ADL. If Grade 2 or 3 hand-foot syndrome occurs, administration of capecitabine should be interrupted until the event resolves or decreases in intensity to Grade 1. Following Grade 3 hand-foot syndrome, subsequent doses of capecitabine should be decreased.

Capecitabine can induce hyperbilirubinemia. Administration of capecitabine should be interrupted if treatment-related elevations in bilirubin of >  $3.0 \times ULN$  or treatment-related elevations in hepatic aminotransferases (ALT, AST) of >  $2.5 \times ULN$  occur. Treatment may be resumed when bilirubin decreases to  $\leq 3.0 \times ULN$  or hepatic aminotransferases decrease to  $\leq 2.5 \times ULN$ /AST) of Grade  $\geq 2$  occur.

# 5.1.3 RISKS ASSOCIATED WITH TRASTUZUMAB EMTANSINE AND CAPECITABINE COMBINATION:

DLTs for the combination of trastuzumab emtansine and capecitabine will be observed during Cycle 1 (Day 1–21) of this study. The combination treatment must be considered as a new treatment during Cycle 1, and no individual dose reduction will be allowed; the general DLT rules will be used instead. Interruptions can be made due to toxicities considered by the investigator to be related to capecitabine. Grade 2–4 toxicities should be interrupted until resolved to Grade 0–1. For Grade 4 toxicities, consideration to discontinue treatment with capecitabine will be made with the adjudication of the SC.

# 5.1.4 DEFINITION OF DOSE **LIMITING** TOXICITY

DLT toxicities will be observed during Cycle 1 (Day 1–21). Please refer to Xeloda<sup>®</sup> SmPC for recommendations on dose reduction.

## **Definition of DLT:**

# **Hematologic**

- Uncomplicated thrombocytopenia Grade 4 which does not recover to ≥ 75-,000/MI before Day 21
- 2. Thrombocytopenia (any grade) complicated with clinically significant bleeding requiring medical intervention such as: platelet transfusion,
cauterization, patients with epistaxis Grade 1 or 2 may have cauterization and this should not be consider as DLT etc.

- 3. Neutropenia Grade 4 lasting > 7 consecutive days
- 4. Febrile neutropenia with an ANC of < 10001,000 cells/mm<sup>3</sup>

#### Non-hematologic

- Diarrhea Grade ≥ 3 which does not decrease to ≤ Grade 2 after 24 hours of starting recommended anti-diarrheal treatment in absence of DPDdeficiency
- 6. Hand-foot syndrome Grade ≥ 3 in absence of DPD deficiency
- 7. Any other treatment-related toxicity ≥ Grade 3 prohibiting the start of the 2nd cycle on dayDay 22 (3 weeks cycle length plus 1 day)

NOTE: If a Grade 2 event requires a dose delay, it will not be considered as DLT. However, if the toxicity does not resolve to Grade 1 or baseline by Day 42, this requires discontinuation and will be considered as DLT.

8. Grade 2 toxicity requiring interruption of treatment for  $> \frac{714}{12}$  days

NOTE: Patients experiencing ≥ Grade 3 hand-foot syndrome or diarrhea or mucositis or Febrile neutropenia with ANC < 500 cells/mm³ during Cycle 1 must be tested for DPD deficiency (central lablaboratory will be appointed). The SC will adjudicate in cases of DLTs that are not covered by the existing DLT criteria.

NOTE TO point 7, if a Grade 2 event requires a dose delay, it will not be considered as DLT.

- 9. Having taken < 14 full doses of capecitabine due to toxicity
- 10. Patient not able to receive 100% of the dose level going into Cycle 2, Day 1

#### 5.1.5 MANAGEMENT OF SPECIFIC ADVERSE EVENTS

#### 5.1.5.1 Trastuzumab Emtansine **Dosage Dose** Modification

Patients should be assessed for toxicity prior to each dose; dosing will occur only if the clinical assessment and laboratory test values are acceptable.

Dose delays and reductions are designed to maximize treatment for those who derive clinical benefit from treatment while ensuring patient safety. Dose delays for trastuzumab emtansine-related toxicity other than those specified below (i.e., infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, cardiotoxicity, and ILD or pneumonitis) are as follows:

Dose delays for trastuzumab emtansine related toxicity other than the onesspecified below (i.e., infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, and cardiotoxicity) are as follows:

• If significant trastuzumab emtansine—related toxicities (other than infusion reactions, thrombocytopenia, hepatotoxicity, neurotoxicity, and cardiotoxicity) have not recovered to Grade 1 or baseline, the next

- scheduled dose may be delayed for up to 42 days from the last dose received. "Significant" and "related" will be based on the judgment of the investigator (in consultation with the Sponsor's Medical Monitor or designee when appropriate). For example, alopecia even if considered related would most likely not be considered to be significant. Fatigue may or may not be considered either related or significant.
- In general, when the significant and related toxicity (or any other toxicity that the investigator chooses to delay dosing for) resolves to Grade 1 or baseline, the patient may resume trastuzumab emtansine if the delay has not exceeded 42 days from the last received dose. Patients should be reevaluated re-evaluated qw during the delay, whenever possible. If dosing resumes, the patient may receive trastuzumab emtansine either at the same dose level as before or at one dose level lower than the previous dose (see Table 2 and Table 3), at the discretion of the investigator. Subsequent cycles should remain the same (q3w or qw), and patients should be assessed for toxicity.
- If a patient requires a dose reduction, dosing will be reduced by one dose level, per Table 2 or Table 3. No dose re-escalation will be allowed.
- If toxicity does not resolve within 42 days from the last dose received, the
  patient will be discontinued from study treatment and will be followed for
  disease progression and survival outcome as described in Section 5.5.
- Patients who experience a Grade 3 or 4 hematologic event should be checked at least <u>qwweekly</u> for recovery. If values do not recover to baseline or Grade ≤ 1 within 42 days from the last dose received, the patient will be discontinued from study treatment.

Table 2 Dose Reductions Reduction for Trastuzumab Emtansine (mBC (Patients with mBC)

| Dose Level | q3w Schedule |
|---------------------------------------------|---------------------|
| 0 | 3.6 mg/kg |
| - 1 | 3.0 mg/kg |
| - 2 | 2.4 mg/kg |
| Indication for<br>further dose<br>reduction | Off study treatment |

q3w = every 3 weeks

Table 3 Dose Reductions for Trastuzumab Emtansine (mGC (Patients with mGC)

| Dose L | evel | qw Schedule |
|------------------------------|------|-------------------------|
| 0 | | 2.4 mg/kg |
| - 1 | | 2 <mark>.0</mark> mg/kg |
| - 2 | | Off study |
| Indication further reduction | dose | Off study |

qw = weekly

In case of toxicities requiring the discontinuation of T-DM1, the patient will be followed-up until the EOS.

Protocol requirements for specific toxicities are outlined below.

## 5.1.5.1.1 Trastuzumab Emtansine Dose Modification for Thrombocytopenia

Platelet counts should be obtained no less frequently than weekly to evaluate recovery whenever any of the events listed below occurs. If platelet counts do not recover to Grade ≤ 1 within 42 days from the last dose received, the patient will be discontinued from study treatment.

No re-escalation of the trastuzumab emtansine dose is allowed.

Note: although complete blood counts with platelets are required within 72 hours prior to study treatment administration at each cycle, the investigator may monitor platelet counts (or any other laboratory test) more frequently as clinically indicated.

In the event of decreased platelet count to Grade 3 ( $< 50,000/\text{mm}^3$ ), do not administer trastuzumab emtansine until platelet counts recover to Grade 1 ( $\ge 75,000/\text{mm}^3$ ), then treat at the same dose level.

Patients receiving trastuzumab emtansine who experience any of the following events listed below a first Grade 4 thrombocytopenia event may, after—adequate recovery to a platelet count of Grade—≤ ≤ 1 (≥ 75,000/µL), mayor baseline, continue treatment with trastuzumab emtansine at one a dose level reduction of 3 mg/kg in subsequent treatment cycles (see Table 2 and Table 3).

#### **Grade 4 Thrombocytopenia:**

Hold study drug until platelet count qualifies for Grade ≤ 1 (≥ 75,000 µL).

- Platelets < 10,000 cells/mm<sup>3</sup> for any duration
- Platelets ≥ 10,000 cells/mm³ but < 25,000 cells/mm³ for more than 7 days</li>

#### **Grade 3 Thrombocytopenia:**

Hold study drug until platelet count qualifies for Grade ≤ 1 ( ≥ 75,000 µL).


- Trastuzumab emtansine 2.4 mg/mg/week dosing
  - Platelets must be ≥ 75,000 µL on day of treatment.
- Trastuzumab emtansine 3.6 mg/kg/q3w dosing:
  - Platelets must be ≥ 75,000 μL on day of treatment.

#### .Patients on Anticoagulation Therapy:

Hold study drug until platelet count qualifies for Grade ≤ 1 (≥ 75,000 µL).

• For platelet count of Grade ≥ 3 (< 50,000 cells/µL) of any duration

Patients at the 3 mg/kg dose level who experience anya Grade 4 thrombocytopenia event may, after adequate recovery as defined above, continue treatment with trastuzumab emtansine at a dose of 2.4 mg/kg in subsequent treatment cycles. Patients who experience a Grade 4 thrombocytopenia event at the 2.4 mg/kg dose level will be discontinued from study treatment. A dose delay of these toxicities should be reassessed at least qw for recovery up to 42 days from the patient's last dose received is permitted.

#### 5.1.5.1.2 Trastuzumab Emtansine Dose Modification for Hepatotoxicity

Table 4 and

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| | <del>Up to</del><br>1.5 × ULN | -> 1.5 3 × ULN | ≥ 3 10 × ULN | ≥ 10 × ULN |
| T-DM1-<br>action | Treat without-<br>dose reduction-<br>or delay | Hold.ª-dose; reduce one dose level when recovered to Grade ≤ 1. Discontinue bif > 2 × ULN and occurs-concurrent with ALT and/or AST elevation > 3 × ULN | Hold a dose; reduce- one dose level when- recovered to- Grade ≤ 1.— Discontinue b if occurs concurrent with ALT and/or AST elevation > 3 × ULN | <del>Discontinue.</del> |

T DM1 = trastuzumab emtansine; ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient-requiring more than two dose reductions must discontinue study treatment.

- <sup>a</sup> A dose delay of up to 42 days after the last received dose is permitted for patients on a q3w schedule or 28 days for patients on a weekly schedule.
- b—Unless a decision is made to hold then continue trastuzumab emtansine treatment based on the results of further evaluation of the situation and agreement by the investigator and the Sponsor. See also Section 0
- € Within 21 days.

| Grade 2 (> 1.5 to $\leq$ 3 × the ULN) | Grade 3<br>(> 3 to ≤ 10 × the ULN) | Grade 4<br>(> 10 × the ULN) |
|---|---|---|
| Do not administer T-DM1 until total bilirubin recovers to Grade ≤ 1, and then treat at the same dose level | Do not administer T-DM1 until total bilirubin recovers to Grade ≤ 1 and then reduce one dose level | Discontinue T-DM1 |

T-DM1 = trastuzumab emtansine; ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

**Table 5**-describe the dose modification guidelines for increases in serum bilirubin and transaminases, respectively. Patients who develop a Grade 4-serum total bilirubin increase or a Grade 4-

# 5.1.5.1.2.1 Concurrent elevations of ALT-and/or-AST increase and bilirubin meeting Hy's Law laboratory criteria

Regardless of dose level, trastuzumab emtansine must discontinue study treatment be permanently. Patients should be checked assessed at least qw-for the recovery of total bilirubin and/or discontinued in patients with ALT and/or AST. If > 3 × ULN and concurrent increase of total bilirubin to > 2 × ULN. All relevant hepatic laboratory tests performed (including AST, ALT, total bilirubin, alkaline phosphatase, activated partial thromboplastin time [aPTT], INR, and albumin) will be entered into the clinical database.

#### 5.1.5.1.2.2 Nodular regenerative hyperplasia (NRH)

Trastuzumab emtansine must be permanently discontinued in patients who are diagnosed with NRH.

# 5.1.5.1.2.3 Transaminase elevations or bilirubin elevation requiring dose adjustment

Patients who experience a Grade 3 elevation of liver function should be checked twice weekly for the recovery of transaminases and/or total bilirubin. If a patient's transaminases and/or ALT and/or ASTtotal bilirubin do not recover to baseline or Grade ≤ 1 (total bilirubin) or Grade ≤ 2 (ALT and/or AST)as per Table 4 and Table 5, within 42– days after from the patient's last dose received, the patient must discontinue study treatment. Please see Section 0 and Table 4 and

| <br>Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|-------------------------------|---------------|--------------|------------|
| <del>Up to</del><br>1.5 × ULN | → 1.5 3 × ULN | ≥ 3 10 × ULN | ≥ 10 × ULN |

| > <u>3 × ULN</u> > <u>3 × ULN</u> |
|-----------------------------------|
|-----------------------------------|

T DM1 = trastuzumab emtansine; ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

- <sup>a</sup> A dose delay of up to 42 days after the last received dose is permitted for patients on a q3w schedule or 28 days for patients on a weekly schedule.
- b—Unless a decision is made to hold then continue trastuzumab emtansine treatment based on the results of further evaluation of the situation and agreement by the investigator and the Spensor. See also Section 0
- <sup>€</sup>Within 21 days.

| Grade 2 | Grade 3 | Grade 4 |
|---|---|---|
| (> 1.5 to ≤ 3 × the ULN) | (> 3 to ≤ 10 × the ULN) | (> 10 × the ULN) |
| Do not administer T-DM1 until total bilirubin recovers to Grade ≤ 1, and then treat at the same dose level | Do not administer T-DM1 until total bilirubin recovers to Grade ≤ 1 and then reduce one dose level | Discontinue T-DM1 |

T-DM1 = trastuzumab emtansine; ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

Table 5 for further information will be discontinued from study treatment.

No re-escalation of the trastuzumab emtansine dose is—allowed.

Table 4 and Table 5 describe the dose modification guidelines for increases in serum bilirubin and transaminases, respectively.

Table 4 Trastuzumab Emtansine Dose Modification: Total Serum Bilirubin

| | Grade 1 | Grade-2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| | <del>Up to</del><br>1.5 × ULN | → 1.5 3 × ULN | ≥ 3–10 × ULN | ≥ 10 × ULN |
| T-DM1-<br>action | Treat without-<br>dose reduction-<br>or delay | Hold *dose; reduce one dose level when recovered to Grade ≤ 1. Discontinue *b if > 2 × ULN and occursconcurrent *c with ALT and/or AST elevation > 3 × ULN | Hold <sup>a</sup> -dose; reduce-<br>one dose level when-<br>recovered to-<br>Grade ≤ 1.—<br>Discontinue bif occurs-<br>concurrent with ALT-<br>and/or AST elevation-<br>> 3 × ULN | <del>Discontinue.</del> |

T DM1 = trastuzumab emtansine: ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

- <sup>a</sup> A dose delay of up to 42 days after the last received dose is permitted for patients on a q3w schedule or 28 days for patients on a weekly schedule.
- b—Unless a decision is made to hold then continue trastuzumab emtansine treatment based on the results of further evaluation of the situation and agreement by the investigator and the Sponsor. See also Section 0
- €—Within 21 days.

| Grade 2 | Grade 3 | Grade 4 |
|---|---|---|
| (> 1.5 to ≤ 3 × the ULN) | (> 3 to ≤ 10 × the ULN) | (> 10 × the ULN) |
| Do not administer T-DM1 until total bilirubin recovers to Grade ≤ 1, and then treat at the same dose level | Do not administer T-DM1 until total bilirubin recovers to Grade ≤ 1 and then reduce one dose level | Discontinue T-DM1 |

T-DM1 = trastuzumab emtansine; ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

Table 5 Trastuzumab Emtansine Dose Modification: Serum ALT or AST

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| | <del>Up to</del><br>3 × ULN | → 3 5 × ULN | ≥ 5-20 × ULN | ≥ 20 × ULN |
| T-<br>DM1-<br>action | Treat without<br>dose-<br>reduction or<br>delay | Treat without dose- reduction or delay. Discontinue b-if- occurs concurrent c- with total bilirubin- > 2 × ULN or clinical jaundice | Hold <sup>+</sup> dose; reduce one-<br>dose level when recovered<br>to Grade ≤ 2. Discontinue<br><sup>b</sup> if occurs concurrent <sup>c</sup> with<br>total bilirubin > 2 × ULN or-<br>clinical jaundice | Discontinue |

T DM1 = trastuzumab emtansine; ULN -- upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

<sup>←</sup> Within 21 days.

| Grade 2<br>(> 3 to ≤ 5 × the ULN) | Grade 3<br>(> 5 to ≤ 20 × the ULN) | Grade 4 (> 20 × the ULN) |
|---|---|---|
| Treat at the same dose level | Do not administer T-DM1<br>until AST/ALT recovers to<br>Grade ≤ 2, and then<br>reduce one dose level | Discontinue T-DM1 |

ALT = alanine transaminase; AST = aspartate transaminase; T-DM1 = trastuzumab emtansine; ULN = upper limit of normal.

Note: A maximum of two trastuzumab emtansine dose reductions is allowed. A patient requiring more than two dose reductions must discontinue study treatment.

#### 5.1.5.1.3 Trastuzumab Emtansine Dose Modification for Neurotoxicity

DM1, an anti-microtubule agent, can potentially cause peripheral neuropathy. Patients should be examined for signs of peripheral neuropathy prior to each dose of trastuzumab emtansine. Patients who experience Grade ≥ 3 neurotoxicity in the form of peripheral neuropathy that does not resolve to Grade ≤ 2 within 42 days after last dose received will be discontinued from study treatment.

Patients receiving trastuzumab emtansine who experience Grade—3 or 4 peripheral neuropathy that does not resolve to Grade ≤ 2 within 42—days after the last dose received will be discontinued from study—treatment.

<sup>&</sup>lt;sup>a</sup>—A dose delay of up to 42 days after the last received dose is permitted for patients on a q3w schedule or 28 days for patients on a weekly schedule.

b—Unless a decision is made to hold then continue trastuzumab emtansine treatment based on the results of further evaluation of the situation and agreement by the investigator and the Sponsor. See also Section 0

#### 5.1.5.1.4 Trastuzumab Emtansine Dose Modification for Cardiotoxicity

Patients without significant cardiac history and with a baseline LVEF ≥ 50% as determined by ECHO or MUGA scan are eligible for study participation. Ejection fractions will be monitored according to during the schedules last week of Cycle 1, Cycle 3 and every third cycle thereafter until the assessment in Appendix 1-at the safety follow-up visit.

Figure 6 summarizes the management of trastuzumab emtansine on the basis of measured LVEF and changes in LVEF from baseline in patients. If the LVEF is reported as a range, the median of the range should be taken. If an investigator is concerned that an AE may be related to cardiac dysfunction, an additional LVEF measurement may be performed. Trastuzumab emtansine will be discontinued in any patient who develops symptomatic CHF. CHF should be treated and monitored according to standard medical practice.

The decision to stop or continue trastuzumab emtansine should be based on the algorithm shown in Figure 6. Trastuzumab emtansine must be discontinued in all patients for whom a confirmed drop of LVEF to below 40% is documented (with a repeat assessment within 21 days). For patients whose LVEF drops to values between 40% and 45% with an absolute decrease in LVEF of  $\geq$  10% points from baseline, trastuzumab emtansine should be held. For these patients, the LVEF should be repeated in 21 days, and trastuzumab emtansine should be discontinued if the LVEF has not recovered to within 10% absolute difference below baseline. If clinically significant cardiac dysfunction or cardiac failure develops or persists or if significant medical management is required to maintain ejection fraction, the patient should be discontinued from study treatment.

Figure 6 Algorithm for Continuation and Discontinuation of Trastuzumab Emtansine Based on Left Ventricular Ejection Fraction Assessments in Patients



CHF = congestive heart failure; LVEF = left ventricular ejection fraction.

Note: LVEF assessment results must be reviewed before the next scheduled trastuzumab emtansine infusion.

- <sup>a</sup> LVEF can be repeated within 21 days, and trastuzumab emtansine should be discontinued if LVEF < 40% is confirmed. Trastuzumab emtansine should be held while the repeat LVEF is obtained.
- b After a second consecutive confirmatory result, trastuzumab emtansine should be discontinued if the LVEF is confirmed to be ≥ 10% points below baseline or if medical management was required to correct the LVEF.

### 5.1.5.1.5 Trastuzumab Emtansine Dose Modification/Management for Infusion-related Reactions, Hypersensitivity Reactions

No pre-medication for Trastuzumab emtansine treatment should be interrupted in patients with severe infusion-related reactions. Trastuzumab emtansine treatment should be permanently discontinued in the first event of life-threatening infusion-related reactions.

Infusion of trastuzumab emtansine is required; however, pre medication is allowed at should be interrupted for patients who develop dyspnea or clinically significant hypotension.

The infusion should be slowed to ≤ 50% or interrupted for patients who experience any other infusion-related symptoms. When the investigator's discretion. patient's symptoms have completely resolved, the infusion may be continued at ≤ 50% of the rate prior to the reaction and increased in 50% increments every 30 minutes as tolerated. Infusions may be restarted at the full rate during the next cycle.

Patients who experience trastuzumab emtansine infusion-related temperature elevations ofto > 38.5°C and/or other-minor infusion-related symptoms may be treated symptomatically with acetaminophen and/or H1 and H2 receptor antagonists (e.g., diphenhydramine and ranitidine, respectively). hydrochloride. Serious infusion-related events (Grade ≥ 3 allergic reaction or acute respiratory distress syndrome [ARDS]) manifested by dyspnea, hypotension, wheezing, bronchospasm, tachycardia, reduced oxygen saturation, or respiratory distress should be managed with supportive therapies as clinically indicated according to standard clinical practice. Patients who experience a Grade ≥ 3 allergic reaction or ARDS care, such as oxygen, beta agonists, antihistamines, antipyretics, or corticosteroids at the investigator's discretion. Pre-medication with corticosteroids, antihistamines, and antipyretics may be used before subsequent infusions of trastuzumab emtansine at the investigator's discretion. Patients should be monitored until complete resolution of symptoms. In the event of a true hypersensitivity reaction (i.e., if the severity of reaction increases with subsequent infusions), trastuzumab emtansine treatment must be permanently discontinued. Patients who experience a Grade ≥ 3 hypersensitivity reaction or acute respiratory distress syndrome (ARDS) will be discontinued from study treatment. Patients who have infusion related symptoms, such as chills or fever, may have the infusion rate decreased by 50% or interrupted. When symptoms have resolved, the infusion may be restarted at ≤ 50% of the prior rate and increased in 50% increments every 30 minutes as tolerated. Pre medication may be used before subsequent infusions at the investigator's discretion. Patients should be monitored until complete resolution of symptoms. the study.

Patients who experience a severe delayed infusion reaction will be discontinued from study treatment.

# 5.1.5.1.6 Trastuzumab Emtansine Dose Modification for Pulmonary Toxicity

Cases of ILD, including pneumonitis (including severe, life-threatening cases) and some leading to ARDS or fatal outcome have been reported with trastuzumab emtansine. Treatment with trastuzumab emtansine has to be permanently discontinued in patients who are diagnosed with ILD or pneumonitis.

#### 5.1.5.1.7 Trastuzumab Emtansine Dose Modification for Extravasation

During the clinical development of T-DM1, reactions secondary to extravasation have been observed. These reactions were usually mild and comprised of erythema, tenderness, skin irritation, pain or swelling at the infusion site. Although T-DM1 is not considered as a vesicant, close monitoring of the infusion site for possible subcutaneous infiltration during drug administration is recommended.

#### 5.1.5.2 Capecitabine Dosage Modification

#### Phase—I: mBC Patients with mBC

Capecitabine The dose modifications during Phase I will of capecitabine can be performed according modified if considered appropriate by the investigator (please refer to the description in Section , study design Xeloda® SmPC for mBC recommendations).

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued in patients with mBC.

#### Randomized Phase-II: Exploration of Efficacy: and Safety in mBC

During the Randomized Phase—II, part of the study, the dose of capecitabine will be modified as per the Xeloda<sup>®</sup> Investigator's Brochure (or SMPC). SmPC.

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued in patients with mBC.

#### Phase I: mGC Patients with mGC

Capecitabine The dose modifications during Phase I will of capecitabine can be performed according modified if considered appropriate by the investigator (please refer to the description in Section , study design Xeloda® SmPC for mGC recommendations).

In case of toxicities requiring the discontinuation of capecitabine, single-agent trastuzumab emtansine may be continued in patients with mGC.

#### 5.2 SAFETY PARAMETERS AND DEFINITIONS

# 5.2.3 PROTOCOL-DEFINED EVENTS OF SPECIAL INTEREST/NON-SERIOUS EXPEDITED ADVERSE EVENTS

Non-serious AEs of special interestAESIs are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2 for reporting instructions). AEs of special interest AESIs for this study include the following:

Potential <u>Drug</u>drug-induced liver injury

Any potential case of drug-induced liver injury as assessed by laboratory criteria for Hy's Lawlaw will be considered as a protocol-defined event of special interest and will need to be reported to the Sponsor expeditiously. The following laboratory abnormalities define potential Hy's Law cases:

The following laboratory abnormalities define potential Hy's law cases:

AST and/or ALT elevations that are > 3 × the ULN

Concurrent with concurrent elevation (within 21 days of AST and/or ALT elevations) of of total bilirubin > 2 × the ULN, except in patients with documented Gilbert Gilbert's syndrome. For patients with Gilbert's syndrome, elevation of direct bilirubin > 2 × ULN should be used instead

#### Suspected transmission of an infectious agent by the study drug:

• Defined as any organism, virus, or infectious particle (e.g., prion protein transmitting transmissible spongiform encephalopathy), both pathogenic and non-pathogenic. A transmission of an infectious agent may be suspected from clinical symptoms or laboratory findings indicating an infection in a patient exposed to a medicinal product. This term ONLY applies when a contamination of the study drug is suspected, NOT for infections supported by the mode of action, e.g., immunosuppression.

### 5.3 METHODS AND TIMING FOR CAPTURING AND ASSESSING SAFETY PARAMETERS

#### 5.3.1 ADVERSE EVENT REPORTING PERIOD

Investigators will seek information on AEs at each patient contact. All AEs, whether reported by the patient or noted by study personnel, will be recorded in the patient's medical record and on the AE eCRF.

After informed consent has been obtained but prior to initiation of study drug, only SAEs caused by a protocol-mandated intervention should be reported (e.g., SAEs related to invasive procedures such as biopsies, medication washout, or no treatment run-in).

After initiation of study treatment, all AEs, regardless of relationship to study drug, will be reported until 30 days after the last administration of study drug or study discontinuation/termination, whichever is later. After this period, investigators should report any deaths, all SAEs, or other AEs and non-serious AESIs (regardless of concern that are believed causality) occurring to be related to prior a patient after the treatment withof that patient has ended should be reported to the Sponsor if the investigator becomes aware of them. The investigator is not required to actively monitor patients after the study drughas ended (see Section 5.6).

#### 5.3.5 PROCEDURES FOR RECORDING ADVERSE EVENTS

#### 5.3.5.1 Diagnosis **Vv**ersus Signs and Symptoms

#### Infusion-Rrelated Reactions

AEs that occur during or within 24 hours after study drug infusion should be captured as individual signs and symptoms rather than a diagnosis of allergic reaction or infusion-related reaction. However, a diagnosis has to be captured as an AE if signs and symptoms constitute a diagnosis of allergic reaction/hypersensitivity or infusion-related reaction and are classified as SAEs; all such symptoms have to be described in the narrative (e.g., in the Additional Case Details field of the eCRF).

#### 5.6 POST-STUDY ADVERSE EVENTS

At the last scheduled study completion/early termination visit, the investigator should instruct each patient to report to the investigator any subsequent AEs

that the patient's personal physician believes could be related or not related to prior studythe drug treatmentunder observation.

The investigator should notify the Sponsor of any death, SAE or other AE of concernAESI occurring at any time after a patient has discontinued study participation if the event is believed to be related to prior study drug treatment or study procedures. The Sponsor should also be notified if the investigator becomes aware of the development of cancer or a congenital anomaly/birth defect in a subsequently conceived offspring of a patient that participated in this study.

The investigator does not need to actively monitor patients for AEs once the trial has ended. The investigator should report these events to the Sponsor-Safety Risk Management on the AE eCRF. If the AE eCRF is no longer available, the investigator should report the event directly to Roche/Genentech Safety Risk Management via telephone or via phone at +1-888-835-2555 facsimile using the Roche Clinical Trial (SAE) Reporting Form.

# 5.7 EXPEDITED REPORTING TO HEALTH AUTHORITIES, INVESTIGATORS, INSTITUTIONAL REVIEW BOARDS, AND ETHICS COMMITTEES

The Steering Committee iDMC will closely monitor the incidence of these expected events during the study. An aggregate report of any clinically relevant imbalances that do not favor the test product will be submitted to health authorities.

#### 6. <u>STATISTICAL CONSIDERATIONS AND ANALYSIS</u> PLAN

#### Phase—I: mBC Patients with mBC:

Enrollment into Cohort—1, patients with HER2-positive mBC-patients, will open first.

Enrolled patients will receive study drug until Investigator assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician or study termination by the Sponsor.

#### Phase II: Exploration of Efficacy: mBC Patients

Phase II will include only Cohort 1, i.e. mBC patients. Patients in Cohort 1, who achieved MTD level will continue with the Phase II part to be assessed for efficacy and safety. Additional patients will be enrolled in this phase in order to achieve the required sample size for this part of the study.

Enrolled patients will receive study drug until Investigator-assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician, or study termination by the Sponsor.

Randomized Phase II: Exploration of Efficacy and Safety in mBC Patients randomized in Phase II will receive study drug until Investigator-assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician, or study termination by the Sponsor.

The final analysis of Randomized Phase—II part of this study for ORR will be performed at the end of studyEOS (defined in Section 3.2).

#### Phase I: Patients with mGC Patients:

Once MTD is established for Cohort—1, enrollment of patients with HER2-positive and locally advanced or mGC patients—into Cohort—2 will be opened.

Enrolled patients will receive study drug until Investigator-assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician, or study termination by the Sponsor.

#### 6.1 DETERMINATION OF SAMPLE SIZE

#### Sample Size for Phase—I: mBC

This part will be based on a classical 3 byplus 3 Phase—I design. From 3A minimum of 6 and up to 18 patients mightwill be enrolled into Cohort—1. There is no formal sample size estimation for this part.

# Sample Size for Randomized Phase—II: Exploration of Efficacy: and Safety in mBC

Assuming a preferable BORR rate of 75% to 80% in Cohort 1 (mBC patients) and aiming for a precision of 8 10%, lower limit of 95% confidence interval of at least 65%, a total of 100 patients would need to be evaluable for Cohort 1.

Approximately 117 patients (78 patients in the combination of T-DM1 and capecitabine respective 39 patients in TDM1 treatment group), including a 10% withdrawal rate, will be randomized with a 2:1 ratio to the combination of T-DM1 and capecitabine or T-DM1.

Point estimates and 95% Clopper-Pearson exact Cls are tabulated for a range of possible BOR outcomes for both treatment groups in Table 8.

Table 8 Sample Size Based on BOR

| Total number of patients is 100 (Phase II) | |
|---|---|
| Number of Patients/ Response 95% Clopper Pearson Confidence Intervals | |
| 75 patients (75%) | <del>65-83%</del> |
| 80 patients (80%) | <del>71 87%</del> |
| Total number of patients adjusted for 10% withdrawal rate is 110 patients | |

| N (T-DM1 and capecitabine)* = 70 patients* | |
|---|---|
| BOR rate [%] | 95% CI (within the treatment group) [%] |
| 57.5 | (45.1–69.2) |
| 60.0 | (47.6–71.5) |
| 62.5 | (50.1–73.8) |
| 65.0 | (52.7–76.0) |
| 67.5 | (55.2–78.2) |
| N (T-DM1) = 35 patients* | N (T-DM1) = 35 patients* |
| BOR rate [%] | 95% CI (within the treatment group) [%] |
| 37.0 | (21.4–54.9) |
| 40.0 | (23.9–57.9) |
| 43.0 | (23.9–57.9) |
| 43.0 | (26.4–60.8) |
| 43.0<br>46.0 | (26.4–60.8)<br>(29.1–63.6) |
| 43.0<br>46.0<br>49.0 | (26.4–60.8) (29.1–63.6) (31.8–66.4) hout adjustment for withdrawal; CI = confidence |

For example, the observed BOR of 75% could be estimated to be within 65% and 83% with a probability of 95% (Clopper Pearson exact confidence intervals). Adjusting for a withdrawal rate of approximately 10%, 110 patients will be enrolled in this phase. Patients from the Phase I (Cohort 1), who received the same dose of study medication during Phase I as chosen dose during Phase II, will contribute to the sample size of 110 patients.

The BOR rate of 75% was chosen based on previously published data for trastuzumab and capecitabine (Tjulandin et al. 2011).

Expected BOR rate for patients who received trastuzumab emtansine of 43.6% (95% CI: 38.6%–48.6%) was chosen based on previously published data for T-DM1 in patients with unresectable, locally advanced or mBC previously treated with a taxane and trastuzumab (EMILIA study; Verma et al. 2012).

The BOR rates for patients treated with the combination of T-DM1 and capecitabine were chosen based on recent results from other combination studies of T-DM1 plus chemotherapy or trastuzumab plus capecitabine.

Response rates were based on those observed in patients with HER2-positive mBC in a Phase Ib/IIa study (BP22752) that compared the combination of trastuzumab emtansine with docetaxel, with or without pertuzumab (ORR: 76% [95% CI: 53%–92%]), and also in a Phase II study that compared the combination of trastuzumab with docetaxel, with or without capecitabine (ORRs: 72.7% [95% CI: 63.4%–80.8%] and 70.5% [95% CI: 61.2%–78.8%]; Wardley et al., 2010).

Increased BOR rates for the combination treatment compared with single-agent trastuzumab emtansine are in line with previously published results of a randomized Phase III study in patients with locally advanced or mBC treated with the combination of trastuzumab with capecitabine *versus* capecitabine alone (ORR: 48.1% *versus* 27.0%, odds ratio = 2.50, p = 0.0115; von Minckwitz et al., 2009).

The precision for the BOR estimate of the combination of T-DM1 and capecitabine is approximately 12%, e.g. BOR of 60%, 95% CI of (47.6%, 71.5%). Due to the lower sample size of the treatment group T-DM1, the corresponding precision for the BOR estimate is increased to 18%, e.g. BOR of 46%, 95% CI of (29.1%, 63.6%).

The 2:1 randomization ratio will be applied to allow more patients being exposed to the combination of T-DM1 and capecitabine and to enable a more thorough assessment of the corresponding safety profile.

The estimation of sample size was performed by Nquery<sup>®</sup> and SAS<sup>®</sup> programs.

#### **Stratification Factors**

The following stratification factor will be implemented in the Randomized Phase II of the trial:

 Number of prior lines of treatment for metastatic disease (1 or >1; excluding single-agent hormones)

A treatment line is any regimen given to patient from treatment initiation until confirmed disease progression.

#### Sample Size for Phase-I: mGC

This part will be based on a classical 3 byplus 3 Phase—I design. From 3 to 1812 patients might be enrolled into Cohort—2. There is no formal sample size estimation for this part.

#### 6.2 SUMMARIES OF CONDUCT OF STUDY

#### Phase I: mBC Patients with mBC

Due to a small sample size, per-protocol (PP) population will not be defined for the Phase I, Cohort 1, however major protocol violations will be summarized for this phase.

Major protocol violations will be summarized by treatment dosage. A median follow-up will be estimated for Phase I, Cohort 1.

### Randomized Phase—II: Exploration of Efficacy: and Safety in mBC Patients

For the Randomized Phase–II, Cohort 1, part of the study, a PP population will be defined (Section 6.4).

Patient enrollment, duration of follow-up, discontinuation from study treatment and study, and reasons for discontinuation will be summarized by treatment group for all randomized patients. In addition, major protocol violations will be summarized by treatment arm.

#### Phase-I: Patients with mGC Patients

Due to a small sample size, a PP population will not be defined for the Phase–I, Cohort 2, however major protocol violations will be summarized for this phase.

Major protocol violations will be summarized by treatment dosage. A median follow-up will be estimated for Phase I, Cohort 2.

### 6.3 SUMMARIES OF TREATMENT GROUP COMPARABILITY

#### Phase-I: mBC

As Phase—I is the Dose Finding part of the study, there are no treatment group comparisons for this part of the study.

Demographics, medical history, and baseline characteristics will be summarized. Continuous variable variables will be summarized by means of median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range while categorical variables — by the number and percentage of patients infor each category treatment dosage.

#### Randomized Phase-II: Exploration of Efficacy and Safety in mBC

The Randomized Phase II includes only Cohort 1, hence treatment comparability is also not applicable for this part of the study is designed to explore the efficacy and safety of the combination of T-DM1 and capecitabine compared with T-DM1.

Demographics, medical history, and baseline characteristics will be summarized. Continuous variable variables will be summarized by means of median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range while categorical variables — by the number and percentage of patients infor each category treatment group.

#### Phase-I: mGC

As Phase—I is the Dose Finding part of the study, there are no treatment group comparisons for this part of the study.


Demographics, medical history and baseline characteristics will be summarized. Continuous variable will be summarized by means of median, mean, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles and range while categorical variables — by the number and percentage of patients infor each category treatment dosage.

#### 6.4 EFFICACY ANALYSES

#### Phase-I, Cohort 1: mBC

The main analysis population will be the safety population including allpatients who received at least one dose of study medication (trastuzumabemtansine and capecitabine). DLT evaluable population as defined in Section 6.5.

#### Randomized Phase II: Exploration of Efficacy: in mBC

The main analysis population for the efficacy analysis will be the intent-to-treat population (ITT) including), which will include all new patients enrolled in the Randomized Phase—II and patients from Cohort 1 who achieved the MTD levelpart of the study. The PP population will include all ITT patients who have at least one post-baseline tumor assessment during the Phase—II and no major protocol violations, which will be defined in the statistical analysis plan-(SAP).

#### Phase-I, Cohort 2: mGC

The main analysis population will be the safety population including allpatients who received at least one dose of study medication (trastuzumabemtansine and capecitabine). DLT evaluable population as defined in Section 6.5.

#### 6.4.1 PRIMARY EFFICACY ENDPOINT

#### Phase—I: mBC, Cohort 1: Patients with mBC

The primary objectives are reaching the MTD and establishing a safety profile. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination.

ORR, as a main efficacy endpoint, will be assessed via BORRBOR rate. The BOR is defined as the best response recorded from the date when the MTD is achieved of enrollment until disease progression/recurrence (or, death)., withdrawal of consent or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

#### Randomized Phase-II: Exploration of Efficacy: in mBC Patients

The primary efficacy endpoint for the Randomized Phase—II part of the study is the BORORR as assessed by investigators via BOR. The BOR is defined as the best response recorded from the start of this or randomization into the

Phase-II II part of the study and until disease progression/recurrence-(or, death) or for patients who were involved in Phase I of the study: the best response from the date, withdrawal of the MTD reached until disease progression/recurrence or death.consent or EOS, whichever occurs first. To be assigned a status of PR or CR, i.e., to be a responder, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 28 days after the criteria for response are first met, i.e., patients need to have two consecutive assessments of PR or CR. This status will be assessed only for patients with measurable disease at baseline. Patients with non-measurable disease at baseline will be assessed for the time to event endpoints (e.g. PFS, OS, etc).

The emphasis of the exploratory Randomized Phase II part of the study will not be formal statistical hypothesis testing but the estimation of:

- The BOR rate with corresponding 95% CIs for each treatment group. The justification of the sample size is based on considerations regarding the width of 95% CIs for each treatment group estimate (precision of the corresponding estimate).
- The treatment effect (between treatment groups comparison) with corresponding 95% CIs.

The number and proportions of responders and non-responders (based on BOR) together with two sided, 95% Clopper-Pearson confidence intervals Cls will be presented, for each treatment group.

The difference in BOR between treatment groups will be displayed with associated 95% CIs using the Hauck-Anderson approach.

Logistic analysis will be used to assess the influence of the stratification factor and baseline covariates in an exploratory manner.

#### Phase I: mGC, Cohort 2: Patients with mGC

The primary objectives are reaching the MTD and establishing a safety profile. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination.

ORR, as a main efficacy endpoint, will be assessed via BORRBOR rate. The BOR is defined as the best response recorded from the date when the MTD is achieved of enrollment until disease progression/recurrence (or, death)., withdrawal of consent or EOS, whichever occurs first. The number of patients is very small in this part of the study. Therefore, all analyses will be descriptive.

#### 6.4.2 SECONDARY EFFICACY ENDPOINTS

#### Phase-I, Cohort 1: mBC

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### Randomized Phase-II: Exploration of Efficacy: in mBC

The secondary efficacy endpoints for the Randomized Phase-II will be:

- Time to response (TTR)
- Duration of response (DoR)
- Time to progression (TTP)
- Time to treatment failure (TTF)
- Progression free survival (PFS)
- Clinical benefit rate (CBR)
- Overall survival (OS)

TTR is defined as the time from enrollmentrandomization to first documentation of confirmed PR or CR (whichever occurs first). Patients who do not have a confirmed response will be censored at the date of the last tumor assessment.

DoR is defined as the period from the date of initial confirmed PR or CR until the date of PD or death from any cause. Patients with no documented progression after CR or PR will be censored at the last date, at which they are known to have had the CR or PR, respectively. The method for handling censoring is the same as described for the PFS below. Only patients with BOR of CR or PR (i.e., responders) will be included in the analysis of DoR.

For patients with a BOR of CR or PR, TTR is defined as the time from the date of enrollment into Cohort 1 randomization to the date of first CR or PR. The censoring rules will be similar to those of the PFS.

TTP is defined as time from enrollment into Cohort 1randomization to the first occurrence of PD. Patients who have not progressed at the time of study completion (including patients who have died before PD) or who are lost to follow-up are censored at the date of the last tumor assessment.

TTF is defined as time from enrollment into Cohort 1 randomization until TTF, for example, treatment failure, e.g., to disease progression, death, withdrawal due to AE or lablaboratory abnormality, or refusal of treatment. Patients who do not experience any of the above events while on study will be censored on the day of their last tumor assessment. For patients who were already in Phase I, the start date will be date of first study medication that was chosen for Phase II.

PFS is defined as the time from enrolment into Cohort 1 randomization until the first documented progression of disease or death from any cause, whichever occurs first. For patients who were already enrolled in Cohort 1 during Phase 1, the time to PFS will be defined from the start date of study medication that was chosen for Phase II. Patients with no PFS events will be censored at the time of the last evaluable tumor assessment. Patients with no tumor assessment after the baseline visit at the time of Phase—II will be censored at the time of enrolmentenrollment plus 1 day.

Clinical benefit response includes patients whose best (confirmed) responsewas PR or CR or stable disease that lasts at least 6 months.

OS is defined as the time from the date of enrollment into Cohort

1-randomization until the date of death, regardless of the cause of death.—For patients who were already in Phase I, same rule as for PFS will be applied.

Patients who were alive at the time of the analysis will be censored at the date of the last follow-up assessment.

Estimates for the survivor function of both treatment groups for the time to event variable such as TTR, DoR, TTP, TTF, PFS, and OS, will be obtained by using the Kaplan-Meier approach method. HRs and associated 95% CIs will be estimated from non-stratified and stratified (based on the stratification factor) Cox regression models.

Clinical benefit response includes patients whose best (confirmed) response was PR, CR or SD that lasted at least 6 months. CBR will be summarized in a similar way to the primary efficacy endpoint, ORR as assessed by BOR.

#### Phase-I, Cohort 2: mGC

Due to the small number of patients and the design of this part of the study, no secondary efficacy endpoints will be investigated.

#### 6.5 SAFETY ANALYSES

#### Safety Population Phase-I, Cohort 1: mBC

The DLT evaluable population is defined for all enrolled and treated patients who have not experienced any major protocol violation (including violation of the inclusion and exclusion criteria) and completed Cycle 1.

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

The safety population (SP) Phase I, mBC will include all patients who received at least one dose of study medication during Phase I. Safety endpoints will be summarized for this part of the study and presented by treatment dosage.

Safety parameters will be analysed analyzed in a similar way to safety parameters in Phase–I, Cohort 2: mGC.

#### Randomized Phase-II: Exploration of Efficacy: Safety in mBC

The SP-Phase II, mBC will include all patients who received at least one dose of study medication during the Randomized Phase II part of the study. Safety endpoints will be summarized for this part of the study and presented.by treatment group.

Safety endpoints during Phase–II will be assessed via÷ total AEs, AEs Grade ≥ 3, SAEs, AESIs (as described in Section 5), premature withdrawal from-study and study medication, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.


The incidence of AEs and SAEs will be summarized according to the primary system-organ class (SOC) and within each SOC, by the Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Based on the safety profile of trastuzumab emtansine time to onset of the first episode of any AESI described in Section 5 will also be summarized via Kaplan-Meier estimates. Additional summaries by frequency tables will also be provided for the AESIs. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry, will be presented in shift tables of NCI-CTC grade at baseline *versus* worst grade during treatment for Cohort 1, the Randomized Phase—II and overall part of the study.

LVEF will be summarized over time by means of mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations, will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### Safety Population Phase-I, Cohort 2: mGC

The DLT evaluable population is defined for all enrolled and treated patients who have not experienced any major protocol violation (including violation of the inclusion and exclusion criteria) and have completed Cycle 1.

The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination. The definition of DLTs is presented in Section 5.1.4. DLTs for this part of the study will be summarized by treatment dose.

The SP Phase I, mGC will include all patients who received at least one dose of study medication during Phase I. Safety endpoints will be summarized for this part of the study and presented by treatment dosage.

Safety parameters for this part of the study will be summarized by treatment dose. The summaries of AEs, SAEs, AEs that cause caused discontinuation from the study treatment, and AESIs will be analyzed in a similar way to AEs in Phase-II.

The incidence of AEs and SAEs will be summarized according to the primary system organ class (SOC) and, within each SOC, by MedDRA preferred term. Based on the safety profile of trastuzumab emtansine time to onset of the first episode of any AESI described in Section 5 will also be summarized via Kaplan-Meier estimates. Additional summaries by frequency tables will also be provided for the AESIs. Patients who died will be listed together with the cause of death.

Laboratory parameters, hematology and biochemistry, will be presented in shift tables of NCI-CTC grade at baseline *versus* worst grade during treatment for Phase I, Cohort-2, Phase I and overall.

LVEF will be summarized over time by means of mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

Other safety variables, such as exposure to study medication, concomitant medications and physical examinations will be analyzed in a similar way. The exposure of study medication will be summarized by frequency tables.

ECOG performance status will be summarized over time and the percentage of patients in different categories will be presented by bar charts at different time points.

#### 6.6 PHARMACODYNAMIC ANALYSES

No pharmacodynamic analyses are planned for this study.

#### 6.7 PHARMACOKINETIC ANALYSES

#### For Phase-I only (Patients with mBC and mGC-Patients):

The following PK parameters of trastuzumab emtansine and capecitabine (including but not limited to thesethose listed below) will be determined only in the Phase—I part of the study for Cohort—1 and Cohort—2 in all patients who receive study treatment using either non-compartmental and/or population methods, if data allow:

- Serum concentrations of trastuzumab emtansine (conjugate) and total trastuzumab
- Plasma concentrations of DM1, capecitabine and its active metabolite 5fluorouracil ( 5-FU)
- Total exposure (e.g., AUC)
- Cmax
- Clearance (CL)
- Volume of distribution (V<sub>d</sub>)
- Terminal half life (V<sub>d</sub>
- T<sub>1/2</sub>→

The pharmacokineticsPK of trastuzumab emtansine, total trastuzumab and DM1 will be compared with historical single—agent PK data to evaluate the potential effect of capecitabine on the PK of trastuzumab emtansine and related analytes. The PK of capecitabine and its active metabolite 5-FU in cycleCycle 1 (in the absence of trastuzumab emtansine) will be compared with the PK of cycleCycle 2 (in the presence of trastuzumab emtansine) to evaluate the potential effect of trastuzumab emtansine on the PK of capecitabine and 5-FU.

All PK parameters will be listed and tabulated by treatment dose and by Cohort. Descriptive summary statistics including arithmetic mean, geometric mean (e.g., AUC and C<sub>max</sub>), median, range, SDs.d., and coefficient of variation will be presented for each cohort. Nonlinear mixed effects modeling will be also used but details will be presented in the statistical analysis planSAP.

PK samples can be obtained ad hoc in case of SAE or unexpected toxicities which may suggest a potential drug-drug interaction.

#### 6.8 EXPLORATORY ANALYSES

For all patients a retrospective central confirmation of the HER2 status will be done. Further exploratory analysis for HER2-positive patients— (based on central confirmation) will be done for selected endpoints such as BOR and safety endpoints (AEs, SAEs, AEs with Grade ≥ 3 and AESIs).

For the Randomized Phase—II: Exploration of Efficacy and Safety in mBC Patients with mBC only:

Subgroup analysis for BOR, safety endpoints (AEs, SAEs and AE, AEs with Grade ≥ 3 and AESIs) in Phase II will be presented for: elderly *versus* younger patients, and patients with ECOG 0–1 *versus* ECOG 2. More details about subgroups will be provideded in the statistical analysis plan.

More details about subgroups will be provided in the SAP.

#### Pharmacoeconomic Endpoint:

The resource expenditure due to hospitalizations that are not study-defined evaluations while on study treatment will be evaluated. The number of hospital visits, number of days admitted, and type of visits (emergency department *versus* inpatient care) will be collected. The reason for admission (disease progression *versus* AE) will also be assessed.

#### 6.9 INTERIM ANALYSES

There is no formal efficacy interim analysis.

However, an IDMC will advise whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 20 and 60 patients have received at least 3 cycles (Cycle 3 Day 1) of treatment in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the course of the Randomized Phase II of the study or as requested.

Efficacy data will only be provided if required by the IDMC to estimate the riskbenefit balance for the patients. Further details on the function and logistics of the IDMC will be provided in the IDMC Charter.

The design of this study includes: Phase–I, Randomized Phase–II and different cohorts. Corresponding analyses as described in the protocol will be performed when all data for particular cohort and study phase are collected and cleaned.

# 9. <u>STUDY DOCUMENTATION, MONITORING, AND ADMINISTRATION</u>

#### 9.3 ADMINISTRATIVE STRUCTURE

The study will have a Steering CommitteeSC, iDMC, central laboratory, IxRS, eCRF, and will be conducted by a contract research organization (CRO) together with the Sponsor.

#### 10. REFERENCES

31. Sawaki A, Ohashi Y, Omuro Y, et al. Efficacy of trastuzumab in Japanese patients with HER2-positive advanced gastric or gastroesophageal junction cancer: a subgroup analysis of the Trastuzumab for Gastric Cancer (ToGA) study. Gastric Cancer 2011; epub ahead of print. DOI: 10.1007/s10120-011-0118-12012; 15:313–22.

{...}

40. Verma S, Miles D, Gianni L, et al. Trastuzumab emtansine for HER2-positive advanced breast cancer. N Engl J Med 2012; 367:1783–91.

{...}

- 44. Wardley A, Anton-Torres A, Pivot X, et al. Trastuzumab plus docetaxel with or without capecitabine in patients with HER2-positive advanced/metastatic breast cancer: first efficacy results from the Phase–II MO16419 (CHAT) Study. SABCS 2006; Abstract# 2063.
- 45. Wardley A, Pivot X, Morales-Vasquez F, et al. Randomized phase II trial of first-line trastuzumab plus docetaxel and capecitabine compared with trastuzumab plus docetaxel in HER2-positive metastatic breast cancer. J Clin Oncol. 2010; 28:976-83.
- 46. World Health Organization, World Health Statistics 2011-; http://www.who.int/whosis/whostat/2011/en/

# Appendix 1 Schedule of Assessments

Table 1 Schedule of assessments for mBC patients (Phase-I-and II, Cohort-1 1 and Randomized Phase II)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | onw | Cycle 4<br><del>/ards</del> Onw | <mark>ards</mark> | Safety<br>Follow-Up<br>Visit | Safety<br>Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every <mark>3-</mark> 6<br>months |
| Informed Consent | Xª | | | | | | | | | | | |
| HER2 Status | Xp | | | | | | | | | | | |
| Medical History and Demographics | Х | | | | | | | | | | | |
| Complete Physical Examination | X | | | | | | | | | | | |
| Limited Physical Examination <sup>c</sup> | | Х | | | Х | | | Х | | | Х | |
| Height and Weight <sup>d</sup> | Х | Х | | | Х | | | Х | | | Х | |
| Vital Signs <sup>e</sup> | Х | Х | | | Х | | | Х | | | Х | |
| ECOG Performance Status | Х | Х | | | Х | | | Х | | | Х | |
| Concomitant Medication Reporting | Xf | Х | | | | | Ongoir | ng | | | | |
| Adverse EventAE Reporting | Xa | | | | | Ongoing | | | | | Х | —X <sup>h</sup> |
| 12-lead ECG | Х | | | | | | | | | | | |
| ECHO/MUGA <sup>i</sup> | Xi | | | X <sup>i</sup> — | | | Xi | | | Xi | X <sup>i</sup> — | |
| Tumor Assessments <sup>j</sup> | х | At eyeleCycle 3 (9 weeks after C1 D1randomization), and then every 4 <sup>th</sup> cycle (12 weeks there after thereafter, regardless of dose delay or early discontinuation, until disease progression or study termination) | | | | | х | х | | | | |
| Brain CT or MRI <sup>k</sup> | Х | At the discretion of the investigator, if clinically indicated, until disease progression | | | | | • | | | | | |
| Bone Scan/Imaging <sup>l</sup> | Х | As clinically indicated | | | | | | | | | | |

Table 1 Schedule of assessments for mBC patients (Phase I, Cohort 1 and Randomized Phase II) (cont.)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | | Cycle 4<br><del>ards<mark>Onwa</mark></del> | ırds | Safety<br>Follow-Up<br>Visit | Safety<br>Follow-Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every <mark>3-</mark> 6<br>months |
| Hematology <sup>m</sup> | X | Xn | Xn | Xn | Xn | Xn | Xn | Xn | | | Х | |
| Biochemistryº | Х | X <sup>n</sup> | X <sup>n</sup> | Xn | X <sup>n</sup> | X <sup>n</sup> | Xn | Xn | | | Х | |
| Urinalysis <sup>p</sup> | X | | As clinically indicated | | | | | | Х | | | |
| INR/aPTT | Х | F | As clinically indicated, e.g. for patients receiving anticoagulation therapy | | | | | Х | | | | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Χq | | | Χq | Х | Х |
| PK/PD Samples (see Appendix 2) <sup>r</sup> | | Xr | | | Xr | | | | | | | |
| Assessment of Patient<br>Hospitalizations and/or Hospital<br>Visits | | х | | | Х | | | Х | | | х | |
| Administration of <del>trastuzumab</del> -<br>emtansine <mark>Trastuzumab Emtansine</mark> | | D 2 <sup>s</sup> | | | D 1 <sup>s</sup> | | | D 1 <sup>s</sup> | | | | |
| Administration of capecitabine Capecitabine | | D 1–14 D 1–14 | | | | | | | | | | |
| Overall <del>survival</del> Survival | Х | X | | | | | Х | Х | | | | |
| Randomization into the Phase II<br>Part of the Study | <mark>X</mark> t | | | | | | | | | | | |

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

- 1. NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within **14 days** prior to first treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1).
- 2. All patients will be followed—up every 6 months (except for pregnancy—every, which is at 3 and 6 months) after safety follow-up visit until disease progression progresses for tumor assessment or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than disease progression will continue to undergo tumor assessments every 3—6 months.
- a) Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests. Patients who are on the MTD dose established in Cohort 1 must re consent to be enrolled into Phase II.
- b) HER2-positivity is defined as IHC 3+ or gene amplification by ISH. It will be performed locally for mBC-patients with mBC c)Limited symptom-directed physical examination.
- d) Height to be obtained at screening or at Cycle 1 Day 1 only.
- e) Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f) Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to first study treatment.
- g) During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h) Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatment-related AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i) Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, and on Day 15-21 of Cycle 1, Cycle 3 and every third cycle thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

- j) Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than disease progression PD, continued tumor assessments according to the protocol schedule of assessments is required every 3–6 months.
- a) Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 4 months) as detailed in Section 04.5.1.4 of the protocol and in . A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- k)An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc 99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- I) An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- m) Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and white blood cells (WBC) with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils.
- n) Assessments should be performed at screening, on Day 1, 8 and 15 of Cycles 1–3, on Day 1 of all subsequent cycles, and weekly following any hematologic AE. If capecitabine is discontinued due to toxicity, assessments should be performed weekly (minimum) until resolution of the AE (Grade ≤ 1/ baseline), and on Day 1 of subsequent cycles thereafter. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- o) Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, blood urea nitrogen (BUN<del>)/urea,</del>), creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN).
- p) Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.

- q) Serum β-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.
- r) Pharmacokinetic assessments will be performed during the dose finding period Dose Finding part of the study only (see Appendix 2).
- s)Trastuzumab emtansine will be administered on Day 1 of each 3-weekly cycle for all mBC patients with mBC in Cohort-1 and Randomized Phase-II period of the study except in the first cycle where trastzumabtrastuzumab emtansine will be given on DAYDay 2 (to allow PK sampling).
- t) Patients will be randomized only in the Randomized Phase II part of the study. No blinding will be used, as this is an open-label study. A 2:1 randomization ratio will be applied to allow more patients to be exposed to the combination of T-DM1 and capecitabine, and to enable a more thorough assessment of the corresponding safety profile.

# Appendix 2 Pharmacokinetic Sampling for Phase–I, Metastatic Breast and Gastric Cancer Patients

| | Trastuzumab<br>emtansine, (T-DM1),<br>total trastuzumab and<br>DM1DM1 <sup>a</sup> PK samples | Capecitabine and 5-FU<br>PK samples |
|---|---|---|
| Cycle 1 Day 1 | | |
| Pre-capecitabine dose | | х |
| 30 min post capecitabine dosing | | х |
| 60 min post capecitabine dosing | | х |
| 1.5 hours post capecitabine dosing | | х |
| 2 hours post capecitabine dosing | | х |
| 2.5 hours post capecitabine dosing | | х |
| 4 hours post capecitabine dosing | | x |
| 6 hours post capecitabine dosing | | х |
| Cycle 1 Day 2 | | |
| Pre trastzumab emtansine-T-DM1 dose | x | |
| 15-30 minutesmin after end of trastuzumab emtansine infusion T-DM1infusion | x | |
| Cycle 2 Day 1 | | |
| Pre trastuzumab emtansine or -<br>capecitabine dose | * | x |
| 30 min post capecitabine dosing | | X |
| 60 min 2 hours post capecitabine dosing | | х |
| 4.56 hours post capecitabine dosing | | х |
| Cycle 1 Day 3 | | |
| 24 hours (± 2 hours) after the end of infusion of T-DM1 | × | |
| Cycle 1 Day 8 | | |
| 7 days (± 1 day) after the end of infusion of T-DM1 <sup>a</sup> | × | |
| Cycle 2 Day 1 | | |
| Pre- capecitabine and T-DM1 dose <sup>a</sup> | × | |

| 15–30 min after end of trastuzumab emtansine infusion | x | |
|---|---|---|
| 30 min post capecitabine dosing | | <mark>x</mark> |
| 60 min post capecitabine dosing | | <mark>x</mark> |
| 1.5 hours post capecitabine dosing | | × |
| 2 hours post capecitabine dosing | | х |
| 2.5 hours post capecitabine dosing | | х |
| 4 hours post capecitabine dosing | | х |
| 6 hours post capecitabine dosing | | × |
| Cycle 2 Day 2 | | |
| 24 hours (± 2 hours) after the end of infusion of T-DM1 | × | |
| Cycle 2 Day 7 | | |
| 7 days (± 1 day) after the end of infusion of T-DM1 <sup>a</sup> | × | |
| Cycle 3 | | |
| Pre T-DM1 dose | × | |

PK = pharmacokinetic; 5-FU = 5-fluoruracil

Data from historic studies have determined that results are the lower limit of quantitation.

<sup>&</sup>lt;sup>a</sup> = Plasma DM1 samples will not be collected at Day 7 post-infusion of T-DM1 neither at pre-dose of Cycle 2 and Cycle 3.

# Appendix 6 ECOG Performance Status

| | Scale |
|---|---|
| <mark>Grade</mark> | |
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory |
| | and able to carry out work of a light or sedentary nature, i.e., light housework, office work |
| 2 | Ambulatory and capable of all self-care but unable to |
| | carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair |
| <u>5</u> | Dead |

http://www.ecog.org/general/perf\_stat.html

TITLE:

#### PROTOCOL AMENDMENT ACCEPTANCE FORM

TRASTUZUMAB EMTANSINE (T-DM1) AND
CAPECITABINE FOLLOWED BY A RANDOMIZED,
OPEN-LABEL PHASE II STUDY OF T-DM1 AND
CAPECITABINE VERSUS T-DM1 ALONE IN HER2-

CAPECITABINE VERSUS T-DM1 ALONE IN HER2
POSITIVE METASTATIC BREAST CANCER AND
HER2-POSITIVE LOCALLY ADVANCED OR
METASTATIC GASTRIC CANCER PATIENTS

PHASE I STUDY OF THE COMBINATION OF

PROTOCOL NUMBER: MO28230

**EUDRACT NUMBER:** 2012-001547-46 **IND NUMBER** To be determined


MEDICAL MONITOR: MD

I agree to conduct the study in accordance with the current protocol.

Principal Investigator's Name (print)

Principal Investigator's Signature

Date

F. Hoffmann-La Roche Ltd

Please return the signed original of this form {as instructed by XX [e.g., your local study monitor, the CRO]} [or] {to the contact provided below}. Please retain a copy for your study files.

{Name} {Address}

SPONSOR:

#### PROTOCOL

TITLE: PHASE I STUDY OF THE COMBINATION OF

TRASTUZUMAB EMTANSINE (T-DM1) AND

CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED/METASTATIC GASTRIC CANCER PATIENTS, FOLLOWED BY A RANDOMIZED,

OPEN-LABEL PHASE II STUDY OF

TRASTUZUMAB EMTANSINE AND CAPECITABINE VERSUS TRASTUZUMAB EMTANSINE ALONE IN HER2-POSITIVE METASTATIC BREAST CANCER

PROTOCOL NUMBER: MO28230

**EUDRACT NUMBER:** 2012-001547-46


MEDICAL MONITOR: MD

SPONSOR: F. Hoffmann-La Roche Ltd

**DATE FINAL:** Version : dd-Mmm-2013

DATE AMENDED: Version: 30-Jun-2014

#### PROTOCOL AMENDMENT APPROVAL


The information contained in this document, especially any unpublished data, is the property of F. Hoffmann-La Roche Ltd (or under its control) and therefore is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Ethics Committee or Institutional Review Board. It is understood that this information will not be disclosed to others without written authorization from Roche except to the extent necessary to obtain informed consent from persons to whom the drug may be administered.

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd Protocol MO28231, Version 3
# PROTOCOL AMENDMENT, VERSION 3 RATIONALE

At the request of the Independent Data Monitoring Committee (IDMC), the design of the trial has been changed to increase the sample size for the randomised Part II Exploration of Efficacy and Safety in metastatic breast cancer (mBC) to provide a more meaningful estimation of efficacy. Following identification of the MTD in Phase I, Cohort 1 in mBC (capecitabine 700 mg/m² bid days 1–14 every 3 weeks [q3w]) in combination with trastuzumab emtansine [T-DM1] 3.6 mg/kg q3w), and the subsequent IDMC recommendation of this Dose Level, the protocol has also been simplified to show this information and remove sections describing Phase I dose de-escalation in the mBC part that are no longer relevant.

Additional information relating to weekly dosing of trastuzumab emtansine in locally recurrent/metastatic gastric cancer has become available from the ongoing adaptive phase II/III GATSBY trial. In October 2013, the IDMC recommended the weekly trastuzumab emtansine regimen in preference to the q3w regimen for further evaluation in the phase III part of the trial.

Further minor changes to the protocol have been made according to the latest clinical information and current recommendations. Specifically, the advice on contraception has been updated in line with the latest Herceptin investigators' brochure. The change in contraception period from 6 to 7 months following the last dose of Herceptin treatment was based on a re-assessment of the half-life of Herceptin across multiple clinical trials and taking a more conservative estimated half-life (up to 38 days). Based on a half-life of up to 38 days, it is expected that Herceptin will have cleared from the blood by 7 months. The extension of the contraception period from 6 to 7 months following the last dose of Herceptin treatment has been implemented in the Herceptin Investigator Brochure, v.14 and the Herceptin prescribing information. As trastuzumab is a component of trastuzumab emtansine, it is now advised that patients of child-bearing potential should also use effective contraception for at least 7 months after their last trastuzumab emtansine treatment, and that nursing mothers should wait before beginning breastfeeding for at least 7 months following treatment. This update is not based on any safety findings, and the benefit-risk assessments for both trastuzumab and trastuzumab emtansine are unchanged.

Additional minor changes have been made to improve clarity and consistency. Deleted text appears in black strikethrough. Substantive new information is marked with yellow highlighting. This amendment represents cumulative changes to the original protocol.

# PROTOCOL AMENDMENT, VERSION 3 SUMMARY OF CHANGES

#### STUDY TITLE

PHASE I STUDY OF THE COMBINATION OF TRASTUZUMAB EMTANSINE (T-DM1) AND CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED-OR-METASTATIC GASTRIC CANCER PATIENTS, FOLLOWED BY A RANDOMIZED, OPEN-LABEL PHASE II STUDY OF T-DM1TRASTUZUMAB EMTANSINE AND CAPECITABINE VERSUS T-DM1TRASTUZUMAB EMTANSINE ALONE IN HER2-POSITIVE METASTATIC BREAST CANCER

#### **SYNOPSIS**

**Study Design** 

**{...}** 

## Phase I: MTD Finding, Cohort 1: mBC

Cohort 1 used will open first with a 3 plus 3 classical design to determine the MTD of capecitabine in combination with trastuzumab emtansine. Initially the study had a dose escalation design, but following the occurrence of two DLTs at Dose Level 1 (750 mg/m² capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine, the study design was adapted and the dose de-escalated to 700 mg/m² capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine. At this Dose Level there were no DLTs and following review of the safety data, . Cohort 1 will enroll patients with HER2 positive mBC. The dose tested of trastuzumab emtansine remains fixed at 3.6 mg/kg every 3 weeks (q3w) and 3 dose levels of capecitabine administered twice daily (bid) on Days 1 to 14 in cycles of 3 weeks will be tested. All patients will be treated until disease progression, intolerable toxicity, withdrawn consent, or death. All patients will be followed up until withdrawn consent, death, or up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first.

## Dose Levels Explored in Phase I, Cohort 1

Dose Level 1: 750 mg/m<sup>2</sup> capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine Dose Level 1: 700 mg/m<sup>2</sup> capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine Dose Level 2: 650 mg/m<sup>2</sup> capecitabine bid + 3.6 mg/kg q3w trastuzumab emtansine The rules for determining the MTD are presented below.

If Dose Level 1 is proved too toxic (dose limiting toxicity [DLT] > 1/3 or > 1/6), the dose will be de escalated to one dose level below (Dose Level 1)

If Dose Level 1 is well tolerated (DLT ≤ 1/6), this dose will be considered the MTD and, following the the Independent Data Monitoring Committee (IDMC) agreement recommended that the study should proceed to will be further explore this Dose Level further d in the Randomized Phase II part of the study. If Dose Level 1 is too toxic (DLT >1/6), the dose will be de escalated to Dose Level 2.

If Dose Level 2 is well tolerated (DLT ≤ 1/6), this dose will be considered the MTD and, following iDMC approval, will be further explored in the Randomized Phase II part of the study. However, if Dose Level 2 is too toxic (DLT > 1/6), the combination may be

## **Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 3

considered unfeasible, recruitment will be closed and neither the Randomized Phase II nor mGC cohort will be opened. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk benefit balance and agreement with the Steering Committee (SC).

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

Phase II will be conducted in mBC patients only. This part of the study will explore the efficacy and safety of the combination treatment of trastuzumab emtansine (T-DM1) and capecitabine, at 700 mg/m² bid (the established recommended MTD), compared with T-DM1 trastuzumab emtansine alone in mBC-patients with mBC.

Once the MTD in Cohort 1 is established, Approximately 210 additional 117 patients with HER2-positive mBC-patients will be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to the Phase II part of the study; however, they will be followed -up until end of study (EOS).

Patients will be treated until disease progression/recurrence, intolerable toxicity, withdrawn consent, or death. If capecitabine needs to be discontinued for any reason, trastuzumab emtansine may continue, and the patient will be followed up until EOS. In case of discontinuation of trastuzumab emtansine, patients will be followed up until EOS.

All patients will be followed up until withdrawn consent, death, or up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first.

#### Phase I: MTD Finding, Cohort 2: LA/mGC

Once the capecitabine MTD dose is established in Cohort 1, Cohort 2 will have open, with a 3 plus 3 classical design and to enroll patients with HER2-positive LA/mGC patients. Trastuzumab emtansine will be administered weekly at the dose of 2.4 mg/kg and capecitabine will start at the MTD dose defined in Cohort 1; capecitabine dose level may be de escalated.

All patients will be treated until disease progression, intolerable toxicity, withdrawn consent, or death. All patients will be followed up until withdrawn consent, death, or up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first. The dose levels for capecitabine will be the same as described in Cohort 1, except for Dose Level 1, which will not be explored in mGC patients. Guidelines for dose escalation and de escalation are as follows: Trastuzumab emtansine will be administered weekly at a dose of 2.4 mg/kg and capecitabine will start at dose level -1 (700 mg/m², the MTD defined in Cohort 1), with de-escalation if required as follows:

If the MTD established in Cohort 1 is defined at Dose Level 1:

- This will be the starting dose in Cohort 2. If Dose Level -1 is well tolerated (DLT in ≤ 1/6 patients), this dose will be established as the MTD for LA/mGC
- De escalation: If Dose Level -1 is not tolerated in Cohort 2 (>(DLT in > 1/6 DLTpatients), de-escalation will be to Dose Level -2.

If the MTD established in Cohort 1 is defined at Dose Level -2:

• This will be the starting dose in Cohort 2. If Dose Level 2 is well tolerated (DLT ≤ 1/6), this dose will be established as the MTD for mGC

• De escalation: if Dose Level 2 is not tolerated in Cohort 2 (> 1/6 DLT), is too toxic, the combination of capecitabine with trastuzumab emtansine 2.4 mg/kg every week willmay be considered not feasible for mGC and Cohort 2 unfeasible in LA/mGC, recruitment will be terminated. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue and the LA/mGC part will be closed. However, this will have no impact on trastuzumab emtansine as a single agent, or with the combination, based on risk benefit balance and agreement with the SCcontinuation of the Randomized Phase II mBC part.

### **Duration of treatment and follow-up**

All patients will be treated until investigator-assessed disease progression, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor. If toxicity is considered by the investigator to be related to only one of the two agents, the non-implicated agent can be continued as single-agent therapy.

All patients will be followed up until withdrawal of consent, death, or for up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first.

#### **Number of Patients**

{...}

Randomized Phase II: Exploration of Efficacy and Safety in mBC

Exploration of efficacy and safety in mBC will be based on 417 approximately 210 randomized patients in total.

Phase I, Cohort 2: LA/mGC

A total of 6 to 12 patients will be enrolled.

#### **Target Population**

Phase I, Cohort 1: mBC

{...}

Before entering the study, patients must have received at least one prior treatment regimen for early or metastatic disease, which includes a chemotherapy agent and trastuzumab either separately or in combination.

#### Randomized Phase II: Exploration of Efficacy and Safety in mBC

{...}

Retrospective central confirmation will be used to censor the efficacy population categorize patients for the Randomized Phase II part of subgroup analyses according to central HER2 testing.

Before entering the study-, patients must have received at least one prior treatment regimen, which includes a chemotherapy agent and trastuzumab either separately or in combination.

{...}

## **Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 3

#### **Inclusion Criteria:**

#### For mBC Patients:

1. Male or female.

{...}

6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 67 months after the last dose of study treatment (see Section 5.2.4 in the protocol).

{...}

- 9. Liver function:
  - Total bilirubin ≤ 1.5 × the upper limit of normal (ULN). or direct bilirubin ≤ 1.5
     × ULN in patients with documented Gilbert's syndrome.
  - b) Serum glutamic oxaloacetic transaminase (SGOT)/aspartate transaminase (AST) and serum glutamic pyruvic transaminase (SGPT)/alanine transaminase (ALT) ≤ 2.5 × the-ULN.
  - c) Alkaline phosphatase ≤ 2.5 ×-the-ULN. In patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × the-ULN.
  - d) Evidence of stable liver function during the month prior to enrollment with liver function tests'-(LFTs) fluctuations not exceeding 2.5 × ULN (for AST, ALT) and 1.5 × ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN.

{...}

12. Life expectancy ≥12 weeks

{...}

15. Tumor block or <del>158</del> slides available for retrospective central confirmation of HER2-positivity (central confirmation not necessary for enrollment).

### For LA/mGC Patients:

1. Male or female

{...}

6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 67 months after the last dose of study treatment (see Section 5.2.4 in the protocol).

{...}

- 9. Liver function:
  - a) Total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤ 1.5 × ULN in patients with documented Gilbert's syndrome.
  - b) SGOT/AST and SGPT/ALT ≤ 2.5 × the ULN.
  - c) Alkaline phosphatase ≤ 2.5 × the ULN. In patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × the ULN.

## **Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 3

d) Evidence of stable liver function during the month prior to enrollment with LFTs fluctuations not exceeding 2.5 × ULN (for AST, ALT) and 1.5 × ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN.

{...}

12. Life expectancy ≥12 weeks

{...}

## **Exclusion Criteria:**

#### For mBC Patients:

{...}

- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogues, such as brivudine.
  - b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption.
  - c) Signs or symptoms suggesting that the patient has dihydropyrimidine dehydrogenase (DPD) deficiency.

{...}

23. No signs and symptoms suggestive that the patient has dihydropyrimidine dehydrogenase (DPD) deficiency.

#### For LA/mGC Patients:

 $\{\ldots\}$ 

- 5. Related capecitabine contraindications:
- a) Treatment with sorivudine or its chemically-related analogues, such as brivudine.
  - b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption.
  - c) Signs or symptoms suggesting that the patient has dihydropyrimidine dehydrogenase (DPD) deficiency.

{...}

22. No signs and symptoms suggestive that the patient has dihydropyrimidine dehydrogenase (DPD) deficiency.

#### Length of Study

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to belast 2 years in total (1 year for DoseMTD Finding and, 1 year for the Phase II Exploration of Efficacy and Safety. All patients in mBC).

#### End of Study

The study will be followed up until withdrawn consent, death or up to a maximum of 2 yearsend after the follow-up period has been completed as defined above. Last patient was randomized in the Phase II part of the study, whichever occurs first. In case Dose

## **Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 3

Level 2|ast visit (LPLV) is too toxic, the study may be terminated prematurely. Patients who, at thatdefined as the last data collection point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as which can be either a clinic visit or a single agent, or with the combination, based on risk benefit balance and agreement with the SC|aboratory sample.

#### **End of Study**

Last patient last visit (LPLV) as per definition is the last data collection point that can be either a clinic visit or a laboratory sample (see above length of study).

In case Dose Level -2 is too toxic in LA/mGC, the LA/mGC cohort may be terminated prematurely. Patients who, at that point, experience response according to RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent or with capecitabine, based on the risk-benefit balance and agreement with the SC.

Randomized Phase II Exploration of Efficacy and Safety in mBC: The primary analysis of best overall response (BOR) rate will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever occurs first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after randomization of the first patient. The EOS analysis (approximately 24 months after the last patient is randomized) will include an updated analysis of BOR, which will be done in a purely exploratory manner.

{...}

#### **Safety Outcome Measures**

- DLT assessment/determination of the MTD of capecitabine when combined with trastuzumab emtansine (Phase I only)
- Incidence, nature, and severity by NCI CTCAE version 4v4.0 of adverse events (AEs), serious adverse events (SAEs), AEs that cause leading to discontinuation from either component of the study treatment, and AEs of special interest (AESIs)
- Fatal cases AEs and their causes of death
- Events to monitor
- Laboratory parameters
- LVEF
- Treatment exposure
- Physical examinations
- Vital signs and ECOG performance status
- Premature withdrawal from study medication and/or study

{...}

#### Statistical Analysis Methods

{...}

There is no formal efficacy interim analysis. However, an independent data monitoring committee (IDMC) will advise whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 20 and 60 patients have

## Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 3

received at least 3 cycles of treatment (Cycle 3 Day 1) in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II of the study or as requested.

Efficacy data will only be provided if required by the IDMC to estimate the risk benefit balance for the patients. Further details on the function and logistics of the IDMC will be provided in the IDMC Charter.

Corresponding analyses as described in the protocol will be performed when all data for from both study phases are collected and cleaned.

Randomized Phase II: The primary analysis of BOR will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever occurs first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after randomization of the first patient. The EOS analysis (approximately 24 months after the last patient is randomized) will include an updated analysis of BOR, which will be done in a purely exploratory manner.

{...}

#### Randomized Phase II: Exploration of Efficacy in mBC

The primary efficacy endpoint for the Phase II part of the study is the ORR, as assessed via the BOR. The rate. BOR is defined as the best response recorded from the start orbetween randomization into the Phase II part of the study and until-disease progression or recurrence, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. To be assigned a status of partial response (PR) or complete response (CR), i.e., to be a responder, changes in tumor measurements must be confirmed by repeated assessments performed no less than 28 days after the response criteria are first met, i.e., patients need to have two consecutive assessments of PR or CR.

The emphasis of the exploratory Randomized Phase II part of the study will not be formal statistical primary hypothesis testing but the estimation of:

Theof interest when comparing ORR – as assessed via BOR rate with corresponding 95% confidence intervals (CIs) for each treatment group. The justification of the sample size is based on considerations regarding the width of 95% CIs for each treatment group estimate (precision of the corresponding estimate).

The treatment effect (- between the two treatment groups comparison) with corresponding 95% Cls., combination of trastuzumab emtansine and capecitabine versus trastuzumab emtansine alone:

- H0:  $\pi_{trastuzumab \ emtansine} = \pi_{trastuzumab \ emtansine} + capecitabine}$  where  $\pi_{trastuzumab \ emtansine}$  is BOR in trastuzumab emtansine alone and  $\pi_{trastuzumab \ emtansine} + capecitabine}$  is BOR in trastuzumab emtansine + capecitabine
- H1: π trastuzumab emtansine ≠ π trastuzumab emtansine + capecitabine

The number and proportions of responders and non-responders (based on BOR) together with the two-sided 9095% Clopper-Pearson confidence intervals (CIs) will be presented for each treatment group. The difference in BOR between treatment groups will be displayed with associated 9095% CIs using the Hauck-Anderson approach and p-value for the Fisher's exact test.

{...}

Estimates for the survivor function of both treatment groups for TTR, DoR, TTP, TTF, PFS and OS will be obtained by using the Kaplan-Meier method. Hazard ratios and associated 9095% Cls will be estimated from non-stratified and stratified (based on the stratification factor) Cox regression models.

{...}

#### Safety Endpoints:

Phase I, Cohort 1: MTD-Finding: mBC

{...}

Safety parameters for this study part will also be summarized by treatment dose. The summaries of AEs, SAEs, AEs that cause discontinuation from the study treatment, and AESIs (as described in Section 5), and events to monitor will be analyzed in a similar way to AEs in Phase II. The summaries will include all patients who received at least one dose of study medication.

{...}

#### Randomized Phase II: Exploration of Safety in mBC

Safety endpoints will be summarized by treatment group.

Safety endpoints during the Randomized Phase II part of the study will be assessed via: total AEs, AEs-Grade ≥ 3 AEs, SAEs, premature withdrawal from study medication, AESIs, events to monitor, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

{...}

#### **Exploratory Analyses**

For all patients with mBC (Phase I, cohort 1; Phase II Exploration of Efficacy and Safety in mBC), a retrospective central confirmation of the HER2 status will be done. Further exploratory analysis for analyses will be done according to centrally confirmed HER2 status positive patients (based on central confirmation) will be done for selected endpoints, e.g. BOR and safety (AEs, SAEs, AEs with Grade ≥ 3 AEs, and AESIs). Subgroup analysis for BOR, safety (AEs, SAEs, AEs with Grade ≥ 3, and AESIs) in the Randomized Phase II part of the study will be presented for both treatment groups with respect to: elderly *versus* younger patients, patients with ECOG 0–1 *versus* ECOG 2; and patients with ≤1 *versus* >1 prior treatment line for metastatic disease. More details will be presented in the SAP.

{...}

#### Sample Size for Randomized Phase II: Exploration of Efficacy and Safety in mBC

The sample size for the primary endpoint BOR is based on a Fisher's exact test with an alpha level of 5% (one-sided), power of 80% and the clinical assumption of a BOR rate of 43% with trastuzumab emtansine alone and 62.5% with the combination of

#### Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 3

trastuzumab emtansine and capecitabine. Approximately 417210 patients (78105) patients in the combination of T DM1 and capecitabine respective 39 patients in T DM1each treatment group), including a 4015% withdrawal rate, will be randomized with a 21:1 ratio to either trastuzumab emtansine alone or the combination of T DM1trastuzumab emtansine and capecitabine-or T DM1.

Point estimates and 95% Clopper Pearson exact CIs are tabulated for a range of possible BOR outcomes for both treatment groups:

Table 1: Sample Size Estimation (2:1 randomization)

| Sample size based on BOR N (T DM1 and capecitabine)* = 70 patients* | |
|---|---|
| <del>57.5</del> | (45.1-69.2) |
| 60.0 | <del>(47.6-71.5)</del> |
| 62.5 | (50.1 73.8) |
| 65.0 | (52.7-76.0) |
| <del>67.5</del> | <del>(55.2-78.2)</del> |
| N (T DM1) = 35 patients | * |
| BOR rate [%] | 95% CI (within treatment group) [%] |
| <del>37.0</del> | <del>(21.4-54.9)</del> |
| 40.0 | (23.9-57.9) |
| 43.0 | <del>(26.4–60.8)</del> |
| 46.0 | <del>(29.1-63.6)</del> |
| 49.0 | (31.8-66.4) |
| <ul> <li>* N = Number of patents</li> <li>interval</li> </ul> | tients without adjustment for withdrawal; CI = confidence |
| N (T DM1 and capecitab | ine) / N (T DM1) = 2 |

Expected BOR rate for patients who received trastuzumab emtansine of 43.6% (95% CI: 38.6% – 48.6%) was chosen based on previously published data for trastuzumab emtansine (see Section 6.1 of the main body of the protocol for reference).

The precision for the BOR estimate of the combination of T DM1 and capecitabine is approximately 12%, e.g. BOR of 60%, 95% Cl of (47.6%, 71.5%). Due to the lower sample size of the treatment group T DM1, the corresponding precision for the BOR estimate is increased to 18%, e.g. BOR of 46%, 95% Cl of (29.1%, 63.6%)

A 2:1 randomization will be applied to allow more patients being exposed to the combination of T DM1 and capecitabine. This will enable a more thorough assessment of the corresponding safety profile.

#### Stratification Factors

The following stratification factor will be implemented in the Randomized Phase II part of the study:

 Number of prior lines of treatment for metastatic disease (≤1 or >1; excluding single-agent hormones).

A treatment line is defined as any treatment regimen given to a patient from treatment initiation until confirmed disease progression.

## Sample Size for Phase I, Cohort 2: MTD-Finding: LA/mGC

This part will be based on a classical 3 plus 3 Phase I design. From Between 3 to and 12 patients might be enrolled in Cohort 2. There is no formal sample size estimation for this part.

#### **Interim analysis**

There is no formal interim analysis of efficacy.

An independent data monitoring committee (IDMC) will recommend whether the Randomized Phase II part of the study can commence.

The IDMC will also monitor safety outcomes after 25, 75, and 150 patients have received at least 3 cycles of treatment (Cycle 3 Day 21) in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II part of the study or as requested.

Efficacy data will be provided only if required by the IDMC to estimate the risk-benefit balance for the patients. Further details on the function and logistics of the IDMC will be provided in the IDMC Charter.

#### **SECTION 1**

# 1.1.1 HER2-Positive Breast Cancer, Metastatic Breast Cancer

Breast cancer (BC) is the most common cancer in women worldwide, both in the developed and the developing world (WHO, World Health Statistics. 2011), world<sup>1</sup>, with approximately an estimated 1.3867 million new cases diagnosed in 20082012. It is also the leading cause of cancer death in females in less developed regions, accounting for 458,400324,000 deaths (14.3% of all cancer deaths) in 2008 (Jemal et al. 2011). Almost 100,000-2012, and the second most common cause of these BC related cancer death in women in more developed regions (198,000 deaths-occurred in patients whose tumors overexpressed human epidermal growth factor receptor 2 (HER2) receptors., 15.4%) after lung cancer. Metastatic breast cancer (mBC) is incurable, with the primary goal of treatment to extend life and palliate symptoms while preserving quality of life.

{...}

However, virtually disease progresses in almost all patients with HER2-positive mBC develop progressive disease (PD) and these patients require additional therapies. Importantly, such tumors continue to express high levels of HER2 (Spector et al. 2005), and neither the process of internalization nor the level of surface expression is altered when HER2 is bound by trastuzumab (Austin et al. 2004). HER2-directed combination therapy beyond progression for HER2-positive mBC is an accepted palliative treatment approach. 8

An accepted example of second line therapy for HER2 positive mBC therapy is lapatinib in combination with capecitabine as a treatment for patients who have received trastuzumab and a taxane for advanced disease. In a After progression, the standard strategy is further HER2-directed therapy, either continuing trastuzumab with a different chemotherapy agent (eg trastuzumab plus capecitabine), or changing to a different HER2-directed regimen (eg lapatinib plus capecitabine). In a randomized Phase III trial, GBG26, in patients whose disease had progressed on previous trastuzumab-containing therapy, the combination of trastuzumab and capecitabine was associated with significantly improved time to progression (TTP) (hazard ratio [HR] 0.69, median 8.2 versus 5.6 months, respectively) and ORR (48% versus 27%) compared with capecitabine alone. In another Phase III trial involving patients with advanced HER2-positive BC previously treated with an anthracycline, a taxane, and trastuzumab, the addition of lapatinib to capecitabine resulted in an increased response rateORR (24% versus 14%) and time to disease progression (TTP (median 6.2 months *versus* 4.3 months) (Geyer et al. 2006), compared with capecitabine alone.9

{...}

# 1.1.2 HER2-Positive Locally Advanced OR METASTATIC GASTRIC CANCER

Gastric cancer (GC) remains one of the most common malignancies in the world with an estimated 989,600952,000 new cases in 2008 (Jemal et al. 2011).2012.1 GC also continues to be a deadly disease; it is the secondthird leading cause of cancer-related death, accounting for 738723,000 deaths (9.78.8% of all cancer deaths) worldwide in 2008 (Ferlay et al. 2010).2012. The only potentially curative treatment for GC is complete resection of localized disease. The overall 5-year survival for all cases, regardless of initial stage at diagnosis, is less than 25% (Catalano et al. 2005; Faivre et al. 1998; Parkin et al. 2005; Power et al. 2010).%.11-14 Among patients with localized disease who undergo curative surgery, approximately 40–60% will have disease recurrence. Patients with unresectable disease due to locally advanced growth or metastatic spread have the poorest prognosis, with an overall 5-year survival rate in the range of 3% to 15% (De Vivo et al. 2000; Ries et al. 2008; Power et al. 2010).%.11,13,14

#### 1.2.1 TRASTUZUMAB EMTANSINE

{...}

Completed and ongoing Phase I and II single-arm studies were conducted to identify the most appropriate dosing regimen for further clinical development, and assess the safety of trastuzumab emtansine have shown clinical activity.

Furthermore, Low levels of DM1 in systemic circulation supported the stability of the linker (Shen et al. ASCPT 2011). The studies also provided an indication of clinical activity and led to randomized Phase II study TDM4450g described in Section 1.2.1.4 showed a significant improvement in PFS with a HR 0.59 (p = 0.0353) and a favorable safety profile. A Phase III study (TDM4370g) is underway comparing evaluation of single-agent trastuzumab emtansine with versus other HER2-targeted directed therapy in combination therapy (capecitabine and lapatinib) for patients with mBC who had received prior with chemotherapy. These trials demonstrated significantly superior PFS and OS with trastuzumab and taxane therapies.emtansine. 26-28

In this study, anthe ORR efwas 25.5% (95% CI: 15.2%–38.5%) was assessed by the investigator; no independent review was performed in this study. The CBR was 39.2% (95% CI: 25.8%–53.1%), and the median PFS was 4.3 months (95% CI: 4.0–6.7).

#### 1.2.1.6 Phase III Study TDM4370g

Roche is conducting A randomized, open-label Phase III trial (TDM4370g) of; EMILIA) compared single-agent trastuzumab emtansine *versus* lapatinib and capecitabine in patients with HER2-positive locally advanced unresectable BC or mBC who havehad received a prior taxane and trastuzumab therapy and havehad documented disease progression. The study is ongoing, enrollment is completed, and 991 patients have been enrolled.PD.<sup>27</sup>

Patients arewere randomized in a 1:1 ratio to trastuzumab emtansine or capecitabine plus lapatinib.

Trastuzumab emtansine is administered at 3.6 mg/kg IV q3w. The control arm treatment is or the combination of oral capecitabine at 1,000 mg/m² as oral doses twice daily (bid) on Days 1–14 of a q3w-cycle plus oral lapatinib 1,250 mg/day given as continuous dosing. Study treatment is discontinued based on disease progression Treatment was continued until PD (as assessed by the investigator), unmanageable toxicity, or study termination by Roche/Genentech.

This study of trastuzumab emtansine, met both primary efficacy endpoints of. PFS by independent review and OS in patients with mBC previously treated with a taxane and trastuzumab (HERCEPTIN).

PFS and OS are investigated as were co-primary endpoints in this study, with PFS based on modified RECIST (Therasse et al. 2000) and conducted by the IRB. An additional tumor assessment of PFS is performed after investigator-documented disease progression. Furthermore ORR, DoR, and CBR are included, on the basis of both investigator and independent review of tumor assessments, as RECIST<sup>34</sup> and assessed by independent review. Key secondary endpoints were ORR, DoR, and CBR, determined both by the investigator and by independent review.

Patients—The study demonstrated statistically significant and clinically meaningful improvements in both PFS and OS for trastuzumab emtansine compared with lapatinib plus capecitabine. Median PFS was 9.6 months in the trastuzumab emtansine arm had a median PFS of 9.6 months—versus 6.4 months for patients in the control arm of lapatinib + capecitabine—(HR = 0.65; 95% CI: 0.55–0.77; p < 0.001, log-rank test). Patients in the trastuzumab emtansine arm had a Median OS of was 30.9 months versus 25.1 months—for patients in the control arm of lapatinib + capecitabine, respectively (HR = 0.68; 95% CI: 0.55–0.85; p < 0.001, log-rank test).

This benefit was supported by consistent improvements in all secondary efficacy endpoints, including investigator-assessed PFS, ORR, time to treatment failure (TTF), and the patient-reported outcome of time to symptom progression. The ORR in the trastuzumab emtansine arm was 43.6% (95% CI: 38.6%–48.6%) compared with 30.8% (95% CI: 26.3%–35.7%) in the control arm (based on 786 evaluable patients). Based on safety data analyzed at the data cut off date, Single-agent trastuzumab emtansine appears to have a favorable overall safety profile compared with lapatinib and capecitabine in mBC. The incidence of Grade  $\geq 3$  AEs in the control arm (56.9%; n = 488) was 278; that of trastuzumab emtansine (40.8%; n = 490) was 200. The rates of SAEs for both arms were similar (control arm 18% *versus* trastuzumab emtansine 15.5%).

It was concluded that overall, there is no concern regarding the clinical safety of trastuzumab emtansine for the patient population that was studied, based on the currently available data (Verma et al. 2012).

Based on the results of this phase III trial, both the Food and Drug Administration (FDA) in the US and the European Medicines Agency (EMA) in Europe approved trastuzumab emtansine for the treatment of HER2-positive mBC previously treated with trastuzumab and a taxane.

## 1.2.1.7 Phase III study TDM4997g

A second open-label randomized Phase III trial (TDM4997g; TH3RESA) compared single-agent trastuzumab emtansine *versus* the investigator's choice of therapy in patients with HER2-positive advanced BC who had previously received two or more HER2-directed regimens in the advanced setting, including trastuzumab and lapatinib, and previous taxane therapy in any setting.<sup>28</sup> A total of 602 patients were randomized in a 2:1 ratio (404 to trastuzumab emtansine and 198 to physician's choice).

After median follow-up of approximately 7 months in both arms, 219 patients (54%) in the trastuzumab emtansine group and 129 (65%) in the physician's choice group had experienced PFS events. PFS was significantly improved with trastuzumab emtansine compared with physician's choice (HR 0.528, p<0.0001; median PFS 6.2 months with trastuzumab emtansine *versus* 3.3 months in the control arm. The HR for OS at the interim analysis was 0.552 (95% CI 0.369–0.826) but the stopping boundary was not crossed.

Grade ≥3 AEs occurred less frequently with trastuzumab emtansine than with physician's choice (32% of natients vs 43%). Grade ≥3 neutropenia, diarrhea

physician's choice (32% of patients vs 43%). Grade ≥3 neutropenia, diarrhea, and febrile neutropenia were less common with trastuzumab emtansine than physician's choice, whereas grade ≥3 thrombocytopenia (5% vs 2%) was more common with trastuzumab emtansine.

{...}

#### 1.2.2 CAPECITABINE

{...}

The activity of capecitabine as single-agent chemotherapy was initially demonstrated in two multicenter Phase II clinical trials (before testing of HER2 status was standard) in patients with locally advanced or mBC after failure of a taxane and an anthracycline-containing chemotherapy regimen or for whom further anthracycline therapy was not indicated. In these trials, a total of 236 patients were treated with capecitabine (1,250 mg/m² bid for 2 weeks followed by 1-week rest period). The ORRs (investigator assessment) were 20% (first trial) and 25% (second trial). The median TTP was 3.1 months and 3.2 months, respectively. Median OS was 12.6 months and 12.3 months, respectively.

The combination of capecitabine and docetaxel was studied as treatment for locally advanced or mBC after failure of anthracycline-containing chemotherapy in a multicenter randomized controlled Phase III clinical trial (SO14999).<sup>40</sup> In this trial, 255 patients were randomized to treatment with capecitabine (1,250 mg/m² bid for 2 weeks followed by a 1-week rest period) and docetaxel (75 mg/m² as a

1-hour IV infusion q3w) and 256 patients were randomized to treatment with docetaxel alone (100 mg/m² as a 1-hour IV infusion q3w). OS was superior in the capecitabine plus docetaxel combination arm (HR 0.775; p = 0.0126). Median OS was 14.5 months (capecitabine plus docetaxel) *versus* 11.5 months (docetaxel alone). The ORR in the all-randomized population (investigator assessment) was 41.6% (capecitabine plus docetaxel) *versus* 29.7% (docetaxel alone; p = 0.0058). TTP was superior in the capecitabine plus docetaxel combination arm (HR 0.652; p < 0.0001). The median TTP was 6.1 months (capecitabine plus docetaxel) *versus* 4.2 months (docetaxel alone).

This trial led to the randomized Phase II CHAT trial evaluating the addition of capecitabine to first-line trastuzumab and docetaxel for locally advanced or metastatic HER2-positive mBC.<sup>41</sup> PFS was significantly improved with the addition of capecitabine (HR 0.72; median 17.9 months *versus* 12.8 months in patients receiving docetaxel and trastuzumab without capecitabine), although there was no difference in ORR (71% *versus* 73%, respectively).

# 1.3 STUDY RATIONALE AND RISK-BENEFIT ASSESSMENT

## 1.3.2 FOR MGC

{...}

In the ToGA study in LA/mGC, trastuzumab exposure was lower than that observed in breast cancer studies. Based on this observation, together with pharmacokinetic results and findings from a Phase I study in mBC, it was considered that a weekly trastuzumab emtansine regimen may provide higher cumulative trastuzumab emtansine exposure than the q3w schedule and was therefore chosen for the Phase I, Cohort 2 part of the present study in LA/mGC. This approach has subsequently been supported by findings from stage I of the adaptive phase II/III BO27952 trial in this setting (see Section ). In October 2013, the IDMC for the BO27952 trial recommended selection of the weekly 2.4 mg/kg regimen for further evaluation in the phase III part of the trial based on pharmacokinetic, safety, and efficacy data available at the time.

{...}

#### **SECTION 3: STUDY DESIGN**

{...}

#### **Duration of Treatment and Patient Follow-up**

<u>LengthDuration</u> of treatment: All patients will be treated until disease progression, intolerable investigator-assessed PD, unacceptable toxicity, (of either or both agents), withdrawal of consent, or death, reasons deemed by the treating physician, or study termination by the Sponsor. If toxicity is considered by the

investigator to be related to only one of the two agents, the non-implicated agent can be continued as single-agent therapy.

If at the time of study closure there are patients whose disease has not progressed and who are still receiving study treatment, they will be offered the possibility to continue treatment by enrolling in an extension study.

<u>Patient follow-up:</u> All patients will be followed up until withdrawnwithdrawal of consent, death, or for up to a maximum of 2 years after the last patient was randomized in the Randomized Phase II part of the study, whichever occurs first.

## **Duration of Study, Database Closure and Data Reporting**

The duration of the study is estimated to be approximately 4 years. Recruitment is estimated to belast 2 years in total (1 year for the Dose-MTD-Finding study in mBC and 1 year for the Phase II Exploration of Efficacy and Safety- in mBC). See Section 3.2 for further details about EOS. The study will end after the follow-up period is completed, as defined above. Last patient last visit (LPLV) is defined as the last data collection point that can be either a clinic visit or a laboratory sample. At that time point, the database will be closed.

In the case that in Cohort 1 the Specifically in Phase I, cohort 2, if dose level -2 is too toxic (> 1/6 of dose-limiting toxicity [DLT]), the combination may be considered unfeasible in LA/mGC, recruitment into the LA/mGC cohort will be closed and neither the Randomized Phase II nor mGC cohort will be opened. See Section 3.1.1.3 for details of treatment continuation if patients who, at that point, experience response as per are still responding to treatment at this time. RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or the combination, based on risk benefit balance and agreement with the Steering Committee (SC).

Data may be reported published/presented publicly at the end of each cohort i.e.g., once the MTD for Cohort 1 for mBC has been defined and the dose for Phase II /Exploration of Efficacy and Safety has been selected. The latest point to write, and after the prespecified analyses for the Randomized Phase II exploration of efficacy and safety in mBC. The Clinical Study Report (CSR) will be finalized/published within 1 year after database closure.

#### **Treatment of Patients after Database Closure**

If at the moment of study closure there are patients who have not progressed and are still receiving study treatment, they will be offered the possibility to continue treatment by enrolling in an extension study.

## **Enrollment into Cohort 1**

Dose MTD-finding in patients with mBC (Phase I)

{...}

If Dose Level -2 is found to be too toxic (DLT > 1/6), the combination may be considered unfeasible, the recruitment will be closed and neither the Randomized Phase II nor mGC cohort will be opened. Patients who, at that point, experience response as per RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk benefit balance and agreement with the SC.

{...}

# 3.1.1.2 Overview of Phase II: Exploration of Efficacy and Safety in Patients with mBC

After review of safety data from Part 1, cohort 1, the IDMC recommended a regimen of capecitabine 700 mg/m² bid days 1–14 in combination with trastuzumab emtansine 3.6 mg/kg q3w for further evaluation. The Phase II This part of the study will explore the efficacy and safety of this recommended regimen the combination treatment of T-DM1 and capecitabine, at the established MTD, compared with T-DM1 trastuzumab emtansine alone in mBC patients with HER2-positive mBC. See Section 3.1.1 for details of duration of treatment.

Once the MTD has been defined to treat patients in Phase II, approximately 117Approximately 210 additional patients with HER2-positive mBC will be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to the Phase II part of the study; however, they will be followed-up until end of study (EOS).

Patients will be treated until disease progression/recurrence, intolerableunacceptable toxicity, withdrawn consent, or death. If capecitabine needs to be discontinued for any reason, trastuzumab emtansine may continue, and the patient will be followed up until EOS. In case of discontinuation of trastuzumab emtansine, at the time of study closure there are will be followed up until EOSwhose disease has not progressed and who are still receiving study treatment, they will be offered the possibility to continue treatment by enrolling in an extension study.

All patients will be followed up until withdrawnwithdrawal of consent, death, or up to a maximum of 2 years after the last patient was randomized in the Phase II part of the study, whichever occurs first.

See Section 3.1.1 for further information.

## 3.1.1.3 Overview of Phase I Design in LA/mGC Patients

### Determination of the MTD in Patients with LA/mGC

Cohort 2 will open when the capecitabine MTD is has been established for Cohort 1 and Cohort 2 will enroll patients with HER2-positive locally advanced and LA/mGC. Trastuzumab emtansine will be administered qw at thea fixed dose of 2.4 mg/kg and capecitabine will be started at 700 mg/m² bid, the MTD defined for patients with mBC in Cohort 1. See Section 3.1.1 for further information.

#### **Enrollment into Cohort 2**

Cohort 2 will open with a 3 plus 3 classical design to investigate the feasibility of combination therapy of capecitabine and trastuzumab emtansine in Cohort 2 (enrolling up to 12 patients with LA/mGC) by de-escalating the dose of . The capecitabine dose will be de-escalated from the starting from dose of 700 mg/m² bid (the MTD determinedrecommended in Cohort 1. In case the MTD was not established or the enrollment was stopped for Cohort 1, enrollment into Cohort 2 will not take place.).

The dose levels for de-escalation of capecitabine will be the same as described for Cohort 1, except for Dose Level 1, which will not be explored in patients with mGC (see also Section 3.3.2.42).

If Dose Level -1 (700 mg/m² bid, the MTD established recommended in cohort 1 is defined at Dose Level -1:

This will be the starting dose in Cohort 2. If Dose Level -1) is well tolerated (DLT in  $\leq$  1/6), this dose will be established as the MTD for LA/mGC.

• De-escalation: If Dose Level -1 is not tolerated in Cohort 2 (>(DLT in>1/3) patients or > 1/6 DLTpatients), de-escalation will be to Dose Level -2.

If the MTD established in Cohort 1 is defined at Dose Level -2:

- This will be the starting dose in Cohort 2. If Dose Level -2 is well tolerated (DLT ≤ 1/6), this dose will be established as the MTD for mGC.
- De-escalation: If Dose Level -2 is not tolerated in Cohort 2 (>(DLT in > 1/6 DLT), the combination will be considered not feasible in LA/mGC and Cohort 2 will be terminated. Patients who, at that pointtime, experience response as peraccording to RECIST v.1.1 will be offered the possibility to continue on trastuzumab emtansine as a single agent, or with the combination, based on risk-benefit balance and agreement with the SC

#### 3.1.1.4 Number of Patients

Overall, it is anticipated that the maximum number of patients enrolled into the study will be approximately 147 patients 240.

{...}

### 3.1.2 STEERING COMMITTEE

A SC has been established for this study. Initially, it is composed of the investigators participating in the Phase I, Cohort 1 part of the study and one medical representative and one statistician of the Sponsor. The study design and DLT has definition have been developed by the SC. See the SC Charter for further information.

The SC will collectively review the status of the ongoing patients in Phase I on a regular basis. the SC will also review in due course all available efficacy data and PK information to ensure that safety information is in the context of risk benefit and that dosing is also related to exposure to the drug.

The SC will adjudicate in casesthe event of DLTs that are not covered by the existing DLT criteria.

#### 3.1.3 INDEPENDENT DATA MONITORING COMMITTEE

An independent data monitoring committee (IDMC) will be established for the Randomized Phase II part of the study. The An IDMC will review the safety outcomes for patients enrolled in Phase I, Cohort 1 and adviserecommend whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 2025, 75, and 60-150 patients have received at least 3 cycles (Cycle 3 Day 121) of treatment in the Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the Randomized Phase II part of the study or as requested.

{...}

## 3.3 RATIONALE FOR STUDY DESIGN

#### 3.3.1 RATIONALE FOR PATIENT GROUP SELECTION

{...}

This study will enroll patients diagnosed with the disease, to which the combination HER2-positive mBC or LA/mGC. Capecitabine is intended.an established chemotherapy for both diseases. In patients with HER2-positive mBC or LA/mGC, anti-HER2 therapy has demonstrated activity. Furthermore, the combination of anti-HER2 agenttherapy and capecitabine has been shown to be efficacious in both mBC (von Minckwitz et al. 2011; Geyer et al. 2006) mBC<sup>9,10</sup> and mGC (Bang et al. 2010), and capecitabine is a standard of care treatment for both diseases. Both diseases LA/mGC. Eligible patients for this study will have been shown to benefit from anti-HER2 treatment; therefore, all patients must be diagnosed with HER2-positive disease. Patients with-incurable mBC and locally advanced or mGC, whose tumors are positive for HER2 overexpression,

represent the patient population eligible for study enrollment or LA/mGC overexpressing HER2.

#### 3.3.1.1 Rationale for Phase I

The study design of 3 plus 3 Phase Idesign is a well-established and well-known method for Phase I studies. PK parameters will be collected and analyzed in order to investigate the PK interaction of the drugs under investigation. Since both agents are administered at efficacious doses, the risk of enrolling patients at the sub-optimal doses is minimal.

Following review of preliminary data from Cohort 1 of this study by the SC for patients enrolled to receive 750 mg/m²-capecitabine, where 2 DLTs were observed in 6 evaluable patients, it was decided not to explore dose levels of capecitabine higher than 750 mg/m². According to the investigator assessment and the SC recommendation, the available evidence shows an acceptable positive risk-benefit in all 7 patients treated at Dose Level 1.

As of 7 August 2013, five patients remain on treatment, with a follow up period of 4 to 8 months. Of the two patients who have discontinued treatment, one patient's disease has progressed, and the other discontinuation was based on the investigator's decision, following the central confirmation, that the patient's disease was HER2-negative. Considering the available safety data for all patients (maximum number of cycles is 12), the combination of capecitabine and T-DM1 is well tolerated, except for increases in transaminases and hand foot syndrome. Dose modifications of T-DM1 and/or capecitabine have allowed those patients to continue on treatment. Of note, no SAE has been reported in 6 patients. Latest tumor response data show 2 patients with PR and 4 patients with SD. Any required dose modifications (dose reductions) are allowed for each individual drug as described in Sections 5.1.5.1 and 5.1.5.2 and are in line with the trastuzumab emtansine Investigator's Brochure and Xeloda®-Summary of Product Characteristics.

The combination of T DM1 and capecitabine will be evaluated with a deescalation study design. Patients who are currently receiving the combination of T DM1 and capecitabine 750 mg/m² can continue to receive the dose as perprotocol until there is no longer evidence of positive risk benefit as per investigator assessment and SC endorsement.

The capecitabine dose evaluated in combination with trastuzumab and docetaxel in the CHAT trial was 950 mg/m² bid. However, retrospective evaluations and post hoc analyses of early dose reduction suggest that lower starting doses of capecitabine offer similar efficacy with better tolerability. Therefore the capecitabine starting dose selected in combination with trastuzumab emtansine for the MTD-Finding Phase I part of the present study was 750 mg/m² bid, taking into account the aim of maintaining the good tolerability of trastuzumab emtansine while benefitting from synergy observed between the two agents in nonclinical studies.

The combination of T-DM1 and capecitabine was evaluated with a de-escalation study design. Following the emergence of two DLTs (grade 3 vomiting, grade 3 elevated AST/ALT) at the starting dose of 750 mg/m² bid (days 1–14 q3w) in combination with trastuzumab emtansine 3.6 mg/kg q3w, a de-escalated dose cohort was opened to evaluate capecitabine 700 mg/m² bid combined with the same dose of trastuzumab emtansine. At this dose no DLTs were observed in the six patients treated, and of note, none of the patients had experienced grade ≥3 AEs in cycles delivered after the DLT evaluation period.<sup>45</sup> Following review of safety data from patients treated at these two dose levels, the IDMC recommended the regimen of capecitabine 700 mg/m² bid combined with trastuzumab emtansine 3.6 mg/kg q3w for the phase II exploration of efficacy and safety.

In the ToGA study in LA/mGC, trastuzumab exposure was lower than that observed in breast cancer studies. A weekly trastuzumab emtansine regimen may provide higher cumulative trastuzumab emtansine exposure than the q3w schedule and was therefore chosen for the Phase I, Cohort 2 part of the present study in LA/mGC. This approach has subsequently been supported by findings from stage I of the adaptive phase II/III BO27952 trial in this setting (see Section ).

#### 3.3.1.2 Rationale for Randomized Phase II

The Randomized Phase II part of the study is designed to explore the efficacy and safety of the combination recommended following the Phase I MTD-Finding phase (trastuzumab emtansine 3.6 mg/kg in combination with capecitabine 700 mg/m²) compared with trastuzumab emtansine alone. provide an estimation of the treatment effect of the combination, at the selected MTD, compared with T-DM1 alone.

The patient data will be stratified by previous anti-cancer treatment (excluding single agent hormones) for the treatment of metastatic disease (1 or >1prior lines of treatment). The stratified data will be compared with data from historical studies of single agent trastuzumab emtansine in similar patient populations. This will allow a more robust evaluation of the added treatment effect of Xeloda® within the combination treatment.

A 2:1 randomization will be applied to allow more patients being exposed to the combination of T DM1 and capecitabine. This will enable a more thorough assessment of the corresponding safety profile.

In addition, it will and provide important information on the longer-term safety of the combination.information.

{...}

#### 3.3.2.2 In Patients with mGC

{...}

In the ongoing randomized adaptive phase II/III BO27952 trial evaluating trastuzumab emtansine versus the investigator's choice of taxane therapy in unrectable LA/mGC, two trastuzumab emtansine regimens were evaluated in stage I: 3.6 mg/kg q3w and 2.4 mg/kg qw . In October 2013, the IDMC for the BO27952 trial recommended selection of the weekly 2.4 mg/kg regimen for further evaluation in the phase III part of the trial based on pharmacokinetic, safety, and efficacy data available at the time. This recommendation provides further support for using the weekly regimen in Phase I, Cohort 2 of the present trial.

{...}

#### 3.3.2.3 Rationale for Duration of Treatment

Treatment will be given until disease progression or unacceptable toxicity investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor (see Section 3.1.1 for full information). As of 1 January 2010, of 237 patients enrolled in studies TDM3569g, TDM4258g, and TDM4374g receiving trastuzumab emtansine at 3.6 mg/kg, approximately 30% have tolerated more than 12 cycles, with 14.8% having received more than 17 cycles. Twenty patients (8.4%) have discontinued trastuzumab emtansine due to AEs and 24 patients (10.1%) required dose reductions in trastuzumab emtansine because of AEs. In the absence of intolerable unacceptable toxicity, patients with mBC are generally treated until disease progression.PD. Further support for treatment until PD comes from the EMILIA randomized phase III trial.<sup>27</sup> Among the 490 patients randomized to trastuzumab-emtansine, only 29 (5.9%) discontinued because of adverse events.

{...}

## 3.3.3 PHARMACOKINETIC SAMPLING RATIONALE

The PK is studied only in the Phase I (MTD-Finding) parts (both cohorts 1 and 2). The PK sampling rationale is to characterize the PK of trastuzumab emtansine, total trastuzumab, and DM1capecitabine and their metabolites, to assess any potential drug-drug interaction when trastuzumab emtansine is given in combination with capecitabine, and to explore potential correlations between drug exposure and measures of both efficacy (ORR) and toxicity (alanine transaminase [ALT]/AST, platelets, etc.), if data allow.

{...}

## 3.4.1.4 Secondary Safety Outcome Measures

{...}

- Premature withdrawal from study medication
- Fatal AEs and their causes
- Abnormal I Laboratory parameters values

{...}

- Vital signs and ECOG performance status
- Premature withdrawal from study medication and/or study

## 3.4.2 RANDOMIZED PHASE II: EXPLORATION OF EFFICACY AND SAFFTY IN MBC

{...}

## 3.4.2.3 Primary Safety Outcome Measure

A primary safety outcome is defined only for Phase I, and will be presented for both treatment groups.

### 3.4.2.4 Secondary Safety Outcome Measures

- Premature withdrawal from study medication
- Fatal AEs and their causes
- Events to monitor
- Laboratory parameters
- Abnormal laboratory values
- LVEF
- Exposure to study medication
- Physical examination
- Vital signs and ECOG performance status
- Premature withdrawal from study medication and/or study

## 3.4.3 Phase I: LA/MGC

## 1.1.1.1 Primary Efficacy Outcome Measure

The main objective for Phase I is to determine the MTD of capecitabine when combined with trastuzumab emtansine. The number and the proportion of

patients with DLTs will be used as the primary measure for the MTD determination and will be summarized for each treatment dosage.

## 1.1.1.2 Secondary Efficacy Outcome Measure

The secondary (efficacy) outcome is ORR, based on BOR rate as peraccording to RECIST v.1.1; based on according to investigator assessment.

### **Primary Safety Outcome Measure**

The primary outcome measure is to establish the MTD. The number and the proportion of patients with DLTs will be used as the primary measure for the MTD determination and will be summarized for each treatment dosage.

## 1.1.1.3 Secondary Safety Outcome Measures

Safety endpoints will be summarized for both treatment phases: Dose Finding and Exploration of Efficacy. Again, the summary of safety endpoints will be presented for each treatment dosage:

- Incidence, nature, and severity of AEs, as peraccording to NCI CTCAE v. 4.0
- Incidence, nature, and severity of SAEs, as peraccording to NCI CTCAE v.
   4.0
- Incidence and nature of AEs equal or higher than Grade ≥3 AEs
- Incidence, nature, and severity of AESIs, as peraccording to NCI CTCAE v.
   4.0
- Fatal cases AEs and their causes of death
- Events to monitor
- Laboratory parameters
- LVEF
- Treatment exposure
- Exposure to study medication
- Concomitant medications and physical examination
- Vital signs and ECOG performance status
- Premature withdrawal from study medication and/or study

#### **SECTION 4: MATERIALS AND METHODS**

### 4.1.3 INCLUSION CRITERIA

#### 4.1.3.1 For Patients with mBC

Patients must meet the following criteria for study entry:

#### 1. Male or female

{...}

6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 67 months after the last dose of study treatment (see Section 5.2.4).

{...}

- 9. Liver function:
  - Total bilirubin ≤ 1.5 × upper limit of normal (ULN) or direct bilirubin ≤1.5
     × ULN in patients with documented Gilbert's syndrome.
  - b) Serum glutamic oxaloacetic transaminase (SGOT)/AST and serum glutamic pyruvic transaminase (SGPT)/ALT ≤ 2.5 × the-ULN
  - c) Alkaline phosphatase ≤ 2.5 × the ULN. In patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × the-ULN
  - d) Evidence of stable liver function during the month prior to enrollment with liver function tests'-(LFTs) fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN

{...}

12. Life expectancy ≥12 weeks

### 4.1.3.2 For Patients with LA/mGC

## 1. Male or female

{...}

6. For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception and to continue its use for the duration of study treatment and for 67 months after the last dose of study treatment (see Section 5.2.4).

{...}

9 Liver function:

- a) Total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤1.5 × ULN in patients with documented Gilbert's syndrome
- b) SGOT/AST and serum glutamic pyruvic transaminase (SGPT)//ALT ≤ 2.5 × the-ULN
- c) Alkaline phosphatase ≤ 2.5 × the-ULN. In patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × the-ULN
- d) Evidence of stable liver function in the month prior to enrollment with LFTs fluctuations not exceeding 2.5 x ULN (for AST, ALT) and 1.5 x ULN (for total bilirubin). Patients with bone metastases: AST and ALT ≤ 5.0 x ULN

#### 4.1.4 EXCLUSION CRITERIA

#### 4.1.4.1 For Patients with mBC

- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogues, such as brivudine
  - b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption
- c) Signs or symptoms suggesting that the patient has DPD deficiency {...}
- 22. Previous radiotherapy for the treatment of unresectable, locally advanced/recurrent or mBC is not allowed if:
  - a) The last fraction of radiotherapy has been administered within 14 days prior to first study drug administration (28 days for patients with radiotherapy to control symptoms of brain metastases, see exclusion criterion 8).
  - b) More than 25% of marrow-bearing bone has been irradiated.
  - c) The patient has not recovered from any resulting Any acute toxicity has not resolved to Grade ≤ 1 prior to before first study drug administration.
- 23. No signs and symptoms suggestive that the patient has dihydropyrimidine dehydrogenase (DPD) deficiency

#### 4.1.4.2 For Patients with LA/mGC

{...}

- 5. Related capecitabine contraindications:
  - Treatment with sorivudine or its chemically-related analogues, such as brivudine

- b) Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
- c) Signs or symptoms suggesting that the patient has DPD deficiency

{...}

8. Brain metastases that are symptomatic, or require any radiation, surgery, or steroid therapy to control their symptoms within 2814 days of before first study drug administration

{...}

22. No signs and symptoms suggestive that the patient has DPD deficiency {...}

## 4.2 METHOD OF TREATMENT ASSIGNMENT

In the Randomized Phase II part of the study, patients will be randomized to receive either the combination of T-DM1 and capecitabine or T-DM1 alone. The 2:1 randomization ratio will be applied to allow more patients being exposed to the combination treatment and to enable a more thorough assessment of the corresponding safety profile. trastuzumab emtansine and capecitabine or trastuzumab emtansine alone.

Patients are stratified according to the number of prior lines of treatment for metastatic disease (≤1 or >1, excluding single-agent therapy).

This is an open-label randomized study; therefore, no blinding will be used.

{...}

#### 4.3.2.2 For Patients with LA/mGC

#### **Trastuzumab Emtansine**

{...}

## Capecitabine

Capecitabine will be administered twice at a day starting dose of 700 mg/m² bid, orally, for 14 days followed by a 7-day rest period at (the dose level that was determined during the Dose Finding part of the study in patients with mBC as the MTD in cohort 1, with de-escalation as described in section 3.1.1.3. Capecitabine tablets should be swallowed with water within 30 minutes after a meal. Capecitabine doses can be delayed for up to 4 hours, while keeping the minimal interval of 8 hours between the doses.

{...}

### 4.5.1.1 Medical History and Demographic Data

Demographic data will include age, sex, and self-reported race/ethnicity (unless not allowed per local regulations).

{...}

## 4.5.1.5 Laboratory Assessments

For Patients with mBC:

{...}

#### **Central Laboratory Assessments:**

 Retrospective HER2 status. Retrospective central confirmation will not impact the treatment decisions or primary endpoint of Phase I, Cohort 1 and will be used to validate efficacy analyses in Phase I and to censor the define subgroups for efficacy population for analyses in the Randomized Phase II part of the study

{...}

## 4.5.2.3 Assessments at Study Completion/Early Termination Visit

Patients may remain on study treatment until disease progression as assessed by the investigator, intolerable-assessed PD, unacceptable toxicity, (of either or until the patient wishes to withdraw fromboth agents), withdrawal of consent, death, reasons deemed by the treating physician, or study treatment termination by the Sponsor. Patients who discontinue study treatment will be followed up until EOS and will be asked to return to the clinic approximately 28–42 days after the last study treatment administration for the safety follow-up visit.

#### 4.5.2.4 Follow-up Assessments

After the Study Treatment Discontinuation Visit, all patients (regardless of reason for discontinuation) will have survival status and anti-cancer therapies recorded and will be followed for all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or dies, or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.

Patients who discontinue study drugs for any reason other than disease progression property or withdrawal of consent (e.g., an AE) will continue to be followed according to the tumor assessment schedule until the development withdrawal of disease progression, consent withdrawal, lost to follow up, death, or beginning of another anti-cancer therapy EOS, whichever occurs first.

After the study treatment completion/early termination visit, AEs should be followed as outlined in Section 5.5 and 5.6.

## **SECTION 5: ASSESSMENT OF SAFETY**

### 5.1.1.3 Hepatotoxicity

Hepatotoxicity, predominantly in the form of asymptomatic increases in the concentrations of serum transaminases (Grade 1–4 transaminitis), has been observed in patients while on treatment with trastuzumab emtansine in clinical trials. Transaminase elevations were generally transient. A cumulative effect of trastuzumab emtansine on transaminases has been observed; The incidence of increased AST was substantially higher than that for ALT. The proportion of patients with Grade 1 or 2 increases in transaminases increased with successive cycles, suggesting a modest cumulative effect of trastuzumab emtansine on transaminases; however, no increase over time in the proportion of Grade 3 abnormalities was observed. Patients with elevated transaminases improved to Grade 1 or normal within 30 days of the last dose of trastuzumab emtansine in the majority of the patients.

Serious hepatobiliary disorders, including nodular regenerative hyperplasia (NRH) of the liver and some resulting in fatal liver failure, have been observed in patients treated with trastuzumab emtansine in clinical trials. Rare cases of severe hepatotoxicity, including death due to drug induced liver injury and associated hepatic encephalopathy, have been observed in patients treated with trastuzumab emtansine. While there is evidence of drug-induced liver toxicity (predominantly in the form of asymptomatic increases in the concentrations of serum transaminases) in patients treated with trastuzumab emtansine, its potential to cause acute severe liver injury with clinically meaningful changes in liver function is unclear as Some of the observed cases of acute liver injury were may have been confounded by comorbidities and/or concomitant medications with known hepatotoxic potential and/or underlying conditions. Liver function should be monitored before initiation of treatment and each trastuzumab emtansine dose. Nevertheless, a contributory role of trastuzumab emtansine in these cases cannot be excluded. Therefore, Acute severe liver injury (Hy's law) remains an important potential risk with trastuzumab emtansine. A Hy's law case has the following components:

- Aminotransferase enzymes (ALT/AST) greater than >3 × ULN with concurrent elevation of serum total bilirubin to >2 × ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)
- No other reason can be found to explain the combination of increased aminetransferases and serum total bilirubin, such as viral hepatitis A, B, or C, pre-existing or acute liver disease, or another drug capable of causing the observed injury.
- The finding should be serious as shown by gross jaundice, clinical disability, need for hospital care, and be at least probably drug-induced (by trastuzumab emtansine)

Trastuzumab emtansine has not been studied in patients with serum transaminases  $> 2.5 \times \text{ULN}$  or total bilirubin  $> 1.5 \times \text{ULN}$  before initiation of treatment. Trastuzumab emtansine treatment in patients with serum transaminases  $> 3 \times \text{ULN}$  and concomitant total bilirubin  $> 2 \times \text{ULN}$  should be permanently discontinued.

Patients must have adequate and stable liver function: hepatic transaminases (AST/ALT) and total bilirubin must be within acceptable range, as defined in the protocol, within 4 weeks prior to the first dose of trastuzumab emtansine. Liver function will be monitored prior to each trastuzumab emtansine dose.

{...}

#### 5.1.2 RISKS ASSOCIATED WITH CAPECITABINE

{...}

Capecitabine can induce severe skin reactions such as Stevens-Johnson syndrome and toxic epidermal necrolysis. Capecitbaine should be permanently discontinued in patients who experience a severe skin reaction during treatment.

# 5.1.3 RISKS ASSOCIATED WITH TRASTUZUMAB EMTANSINE AND CAPECITABINE COMBINATION

The two DLTs observed in Phase I, Cohort 1 (in mBC) were grade 3 vomiting in one patient and grade 3 elevated AST and ALT in one patient (see Section ****). Both patients were treated at dose level 1 (capecitabine 750 mg/m² bid, days 1–14) in combination with trastuzumab emtansine 3.6 mg/kg q3w). During Phase I in LA/mGC, DLTs for the combination of trastuzumab emtansine and capecitabine will be observed during Cycle 1 (Days 1–21) of this study.

{...}

## 5.1.5.2 Capecitabine Dosage Modification

#### Phase I: Patients with mBC

The dose of capecitabine can be modified from Cycle 2 onwards if considered appropriate by the investigator (please refer to the Xeloda® SmPC for recommendations).

{...}

## Phase I: Patients with mGC

The dose of capecitabine can be modified from cycle 2 onwards if considered appropriate by the investigator (please refer to Xeloda® SmPC for recommendations).

{...}

# 5.2.3 PROTOCOL-DEFINED EVENTS OF SPECIAL INTEREST/NON-SERIOUS EXPEDITED ADVERSE EVENTS

Non-serious AESIs are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event (see Section 5.4.2 for reporting instructions) regardless of the attribution of causality. AESIs for this study include the following:

Potential drug-induced liver injury

Any potential case of drug-induced liver injury as assessed by laboratory criteria for Hy's law will be considered as a protocol-defined event of special interest and will need to be reported to the Sponsor expeditiously.

The following laboratory abnormalities define potential Hy's law cases:

AST and/or ALT elevations that are > 3 × ULN with concurrent elevation of total bilirubin > 2 × ULN, (or clinical jaundice if total bilirubin measures are not available), except in patients with documented Gilbert's syndrome. For patients with Gilbert's syndrome, elevation of direct bilirubin > 2 × ULN should be used instead

{...}

## 5.2.4 PREGNANCY AND CONTRACEPTION

ICH M3 guidance requires precautions to be taken to minimize risk to fetus or embryo when including women of childbearing potential in clinical studies. These precautions include the use of highly effective contraceptive measures, excluding pregnancy at baseline (serum test), continued pregnancy monitoring, and continued pregnancy testing for up to 67 months following last dose of study drug (follow-up period based on PK considerations).

{...}

For male patients with a female partner of childbearing potential, cooperation of female partner is required (i.e., use of two forms of contraception as stated above) during the study and for at least 67 months following the last dose of study treatment when a highly effective form of contraception is not appropriate.

Based on PK considerations, contraception must continue for the duration of study treatment and for at least 67 months after the last dose of study treatment.

A female patient or partner of a male patient who becomes pregnant during the study must be instructed to stop taking the study medication and immediately inform the investigator. The investigator should report all pregnancies—within 24 hours to the Sponsor, including the partners of male patients, to the Sponsor within 24 hours. The investigator should counsel the patient/partner, and discuss the risks of continuing with the pregnancy and the possible effects on the fetus. Monitoring of the patient/partner should continue until conclusion of the

pregnancy. Pregnancies occurring up to 67 months after the completion of study medication must also be reported to the investigator. Please refer to Section 5.4.3 for reporting procedures.

It is not known whether trastuzumab or trastuzumab emtansine are excreted in human milk. Maternal IgG is excreted in milk and any of these monoclonal antibodies could harm infant growth and development; therefore, women should be advised to discontinue nursing during trastuzumab emtansine therapy and not to breastfeed for at least 67 months following the last dose of either study drug.

{...}

This is to ensure that the fetus is not exposed to the study medication through vaginal absorption. In addition, sperm or blood donation should not occur for at least 67 months after the last dose of study treatment.

### 5.3.1 ADVERSE EVENT REPORTING PERIOD

{...}

After informed consent has been obtained but prior to initiation of study drug, only SAEs caused by a protocol-mandated intervention should be reported (e.g., SAEs related to invasive procedures such as biopsies, discontinuation of medications washout, or no treatment run in) should be reported (see Section  for instructions for reporting SAEs).

After initiation of study treatment, all AEs, regardless of relationship to study drug, will be reported until 2830 days after the last administration of study drug-or study discontinuation/termination, whichever is later. After this period, all SAEs and non-serious AESIs (regardless of causality) occurring to a patient after the treatment of that patient has ended should be reported to the Sponsor if the investigator becomes aware of them. After this period, the investigator is not required to actively monitor for AEs; however, the Sponsor should be notified if the investigator becomes aware of any poststudy SAEs patients after the study has ended (see Section 5.6).

{...}

## 5.4.3 REPORTING REQUIREMENTS FOR PREGNANCIES

## 5.4.3.1 Pregnancies in Female Patients

Female patients of childbearing potential will be instructed to immediately inform the investigator if they become pregnant during the study or within 67 months after the last dose of study drug. A Pregnancy Report eCRF should be completed by the investigator immediately (i.e., no more than 24 hours) after learning of the pregnancy and submitted via the EDC system. A Pregnancy Report will automatically be generated and sent to the Sponsor Safety Risk Management. Pregnancy should not be recorded on the AE eCRF. The investigator should have the patient discontinue the study drug and discuss with the patient the risks

of the pregnancy and the possible effects on the fetus. Monitoring of the patient should continue until conclusion of the pregnancy.

{...}

## 5.4.3.2 Pregnancies in Female Partners of Male Patients

Male patients will be instructed through the Informed Consent Form to immediately inform the investigator if their partner becomes pregnant during the study or within 67 months after the last dose of study drug.

{...}

## 5.6 POST-STUDY ADVERSE EVENTS

At the time of study completion/early termination visit or study discontinuation, the investigator should instruct each patient to report to the investigator any subsequent AEs that the patient's physician believes could be related or not related to the prior study drug under observation treatment or study procedures.

The investigator should notify the Sponsor of any death, SAE or AESI occurring at any time after a patient has discontinued study participation. The investigator is not required to actively monitor patients for AEs after the end of the AE reporting period (defined as 28 days after the last dose of study drug). However, the Sponsor should be notified if the investigator becomes aware of any death or other SAE occurring after the end of the AE reporting period, regardless of causality. The Sponsor should also be notified if the investigator becomes aware of the development of cancer or a congenital anomaly/birth defect in a subsequently conceived offspring of a patient that participated in this study female patient exposed to study drug or the female partner of a male patient exposed to study drug.

The investigator does not need to actively monitor patients for AEs once the trial has ended. The investigator should report the eventthese events directly to Roche Safety Risk Management via telephone or via facsimile using the Roche Clinical Trial (SAE) Reporting Form.

{...}

# SECTION 6: STATISTICAL CONSIDERATIONS AND ANALYSIS PLAN

The design of this study includes: Phase I, Randomized Phase II and different cohorts. Corresponding analyses as described in the protocol will be performed when all data for a particular cohort and study phase are collected and cleaned.

#### Phase I: Patients with mBC:

Enrollment into Cohort 1, patients with HER2-positive mBC, will open first.

Enrolled patients will receive study drug until Investigator-assessed disease progressionPD, unacceptable toxicities, patient consenttoxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.

Randomized Phase II: Exploration of Efficacy and Safety in mBC Patients randomized in Phase II will receive study drug until Investigator assessed disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician, or study termination by the Sponsor.

Patients randomized in Phase II will receive study drug until investigatorassessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.

The final primary analysis of Randomized Phase II part of this study for ORRBOR will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever comes first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after the randomization of the first patient.

The EOS (defined in Section 3.2).analysis will include an updated analysis of BOR, which will be done in a purely exploratory manner.

#### Phase I: Patients with mGC:

Once the MTD is established for Cohort 1, enrollment of patients with HER2-positive and locally advanced or LA/mGC into Cohort 2 will be opened.

Enrolled patients will receive study drug until investigator-assessed disease progressionPD, unacceptable toxicities, patient consenttoxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.

#### 6.1 DETERMINATION OF SAMPLE SIZE

### Sample Size for Phase I: mBC

This part will be based on a classical 3 plus 3 Phase I design. A minimum of 6 and up to 18 patients will be enrolled into Cohort 1. There is no formal sample size estimation for this part.

## Sample Size for Randomized Phase II: Exploration of Efficacy and Safety in mBC

The sample size for the primary endpoint BOR is based on a Fisher's exact test with an alpha level of 5% (one-sided), 48,49 power of 80% and the clinical assumption of a BOR rate of 43% with trastuzumab emtansine alone and 62.5% with the combination of trastuzumab emtansine and capecitabine. Approximately 117210 patients (78105 patients in the combination of T DM1 and capecitabine respective 39 patients in TDM1each treatment group), including a 1015% withdrawal rate, will be randomized with a 21:1 ratio to trastuzumab emtansine alone or the combination of T DM1 trastuzumab emtansine and capecitabine or T-DM1.

Point estimates and 95% Clopper-Pearson exact Cls are tabulated for a range of possible BOR outcomes for both treatment groups in Table 8.
Table 1 Sample Size Based on BOR

| BOR rate [%] | 95% CI (within the treatment group) [%] |
|---|---|
| <del>57.5</del> | <del>(45.1-69.2)</del> |
| 60.0 | <del>(47.6–71.5)</del> |
| 62.5 | (50.1-73.8) |
| 65.0 | (52.7-76.0) |
| <del>67.5</del> | <del>(55.2–78.2)</del> |
| N (T DM1) = 35 patien | 95% CI (within the treatment group) [%] |
| BOR rate [%] | 95% CI (within the treatment group) [%] |
| BOR rate [%] | 95% CI (within the treatment group) [%] |
| BOR rate [%] | 95% CI (within the treatment group) [%] |
| BOR rate [%]<br>37.0<br>40.0 | 95% CI (within the treatment group) [%] (21.4 54.9) (23.9-57.9) |
| BOR rate [%]<br>37.0<br>40.0<br>43.0 | 95% CI (within the treatment group) [%] (21.4 54.9) (23.9 57.9) (26.4 60.8) |

N (T-DM1 and capecitabine) / N (T-DM1) = 2

Expected BOR rate for patients who received trastuzumab emtansine An expected BOR rate of 43.6% (95% CI: 38.6%–48.6%) for patients receiving trastuzumab emtansine alone was chosen based on previously published data for T-DM1 in patients with unresectable, locally advanced or mBC previously treated with a taxane and trastuzumab (EMILIA study; Verma et al. 2012).).27

{...}

The precision for the BOR estimate of the combination of T DM1 and capecitabine is approximately 12%, e.g. BOR of 60%, 95% Cl of (47.6%, 71.5%). Due to the lower sample size of the treatment group T DM1, the corresponding

precision for the BOR estimate is increased to 18%, e.g. BOR of 46%, 95% Cl of (29.1%, 63.6%).

The 2:1 randomization ratio will be applied to allow more patients being exposed to the combination of T DM1 and capecitabine and to enable a more thorough assessment of the corresponding safety profile.

The estimation of sample size was performed by Nquery<sup>®</sup> and <del>SAS</del>EAST<sup>®</sup> programs.

# Stratification Factors

The following stratification factor will be implemented in the Randomized Phase II of the trialstudy:

 Number of prior lines of treatment for metastatic disease (≤1 or >1; excluding single-agent hormones)

A treatment line is any regimen given to a patient from treatment initiation until confirmed disease progression PD.

{...}

# 6.4.1 PRIMARY EFFICACY ENDPOINT

{...}

# Randomized Phase II: Exploration of Efficacy in mBC

The primary efficacy endpoint for the Randomized Phase II part of the study is the ORR as assessed via BOR. The BOR is defined as the best response recorded from the start or randomization into the Phase II part of the study and until disease progression/recurrencePD, death, withdrawal of consent, start of new anticancer treatment, or EOS, whichever occurs first. To be assigned a status of PR or CR, i.e., to be a responder, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 28 days after the criteria for response are first met, i.e., patients need to have two consecutive assessments of PR or CR.

The emphasis of the exploratory Randomized Phase II part of the study will not be formal statistical primary hypothesis testing but the estimation of:

Theof interest when comparing ORR – as assessed via BOR rate with corresponding 95% CIs for each treatment group. The justification of the sample size is based on considerations regarding the width of 95% CIs for each treatment group estimate (precision of the corresponding estimate).

The treatment effect (<u>between the two</u> treatment groups <del>comparison</del>) with corresponding 95% Cls. (combination of trastuzumab emtansine and capecitabine *versus* trastuzumab emtansine alone) is:

- H0: π<sub>TDM1</sub> = π<sub>trastuzumab</sub> emtansine + capecitabine</sub> where π<sub>trastuzumab</sub> emtansine is BOR in TDM1 and π trastuzumab emtansine + capecitabine is BOR in trastuzumab emtansine + capecitabine
- H1: π trastuzumab emtansine ≠ π trastuzumab emtansine + capecitabine

The number and proportions of responders and non-responders (based on BOR) together with 9095% Clopper-Pearson CIs will be presented for each treatment group.

The difference in BOR between treatment groups will be displayed with associated 9095% CIs using the Hauck-Anderson approach and p-values for the Fisher's exact test.

Logistic analysis will be used to assess the influence of the stratification factor and baseline covariates in an exploratory manner.

The primary analysis of BOR will be performed when 70% of the patients have experienced a PFS event or at the end of the trial, whichever comes first. It is estimated that 70% of patients will have experienced a PFS event approximately 26 months after the randomization of the first patient.

{...}

# 6.4.2 SECONDARY EFFICACY ENDPOINTS

{...}

Estimates for the survivor function of both treatment groups for TTR, DoR, TTP, TTF, and OS will be obtained by using the Kaplan-Meier method. HRs and associated 9095% CIs will be estimated from non-stratified and stratified (based on the stratification factor) Cox regression models.

{...}

# 6.5 SAFETY ANALYSES

{...}

# Randomized Phase II: Exploration of Safety in mBC

Safety endpoints during Phase II will be assessed via total AEs, AEs-Grade ≥3 AEs, SAEs, AESIs (as described in Section 5), fatal AEs and their causes, events to monitor, premature withdrawal from study medication and/or study, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

{...}

**Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 3

# 6.8 EXPLORATORY ANALYSES

{...}

For the Randomized Phase II only: Exploration of Efficacy and Safety in Patients with mBC-only:

Subgroup analysis for BOR, safety endpoints (AEs, SAEs, <del>AEs with Grade ≥ 3 AEs, and AESIs) in Phase II will be presented for: elderly *versus* younger patients, <del>and patients with ECOG 0–1 versus ECOG 2, and patients with ≤ versus >1 prior treatment regimen for metastatic disease.</del></del>

# 6.9 INTERIM ANALYSES

There is no formal efficacy interim analysis.

However, an IDMC will adviserecommend whether the Randomized Phase II part of the study can commence. The IDMC will also monitor safety outcomes after 2025, 75, and 60-150 patients have received at least 3 cycles (Cycle 3 Day 1) of treatment in the Randomized Phase II part of the study. Afterwards, the IDMC will monitor accumulating patient safety data every 6 months during the course of the Randomized Phase II of the study or as requested.

# Appendix 1 Schedule of Assessments

# Table 1 Randomized Phase II)

# Schedule of assessments for mBC patients (Phase I, Cohort 1 and

| | Screening <sup>1</sup> | | Cycle 1 | | 1 | Cycle 2–3 | 3 | Сус | le 4 Onw | ards | Safety<br>Follow-Up<br>Visit | Follow-<br>Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 3-6<br>months |
| Informed Consent | Xa | | | | | | | | | | | |
| HER2 Status | Xp | | | | | | | | | | | |
| Medical History and<br>Demographics | × | | | | | | | | | | | |
| Complete Physical Examination | Х | | | | | | | | | | | |
| Limited Physical Examination <sup>c</sup> | | Χ | | | Х | | | Х | | | Х | |
| Height and Weight <sup>d</sup> | Х | Χ | | | Х | | | Х | | | Х | |
| Vital Signs <sup>e</sup> | X | Χ | | | Х | | | Х | | | Х | |
| ECOG Performance Status | X | Χ | | | Х | | | Х | | | Х | |
| Concomitant Medication Reporting | X <sup>f</sup> | Х | | | | | Ongoi | ng | | | | |
| AE Reporting | Χg | | | | | Ongoing | | | | | Х | $X^h$ |
| 12-lead ECG | X | | | | | | | | | | | |
| ECHO/MUGA <sup>i</sup> | Xi | | | Xi | | | Xi | | | Xi | Xi | |
| Tumor Assessments <sup>j</sup> | Х | | At Cycle 3 (9 weeks after randomization), and then every 4 <sup>th</sup> cycle (12 weeks thereafter, regardless of dose delay or early discontinuation) until <del>disease</del> X progressionPD or study termination), whichever occurs earlier | | | | | | | | | X |
| Brain CT or MRI <sup>k</sup> | Х | | At th | e discretion | on of the i | nvestigate | or, if clinic | ally indica | ated, until | disease | <del>progression<mark>PD</mark></del> | |

| Bone S | Scan/Imaging <sup>l</sup> | Х | As clinically indicated |
|--------|---------------------------|---|-------------------------|
|--------|---------------------------|---|-------------------------|

# Appendix 1 Schedule of Assessments (cont.)

Table 1 Schedule of assessments for mBC patients (Phase I, Cohort 1 and Randomized Phase II) (cont.)

| | Screening <sup>1</sup> | Cycle 1 | | | | Cycle 2–3 | | | e 4 Onwa | ırds | Safety<br>Follow-Up<br>Visit | Follow-<br>Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 3-6<br>months |
| Hematology <sup>m</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | Xn | X <sup>n</sup> | X <sup>n</sup> | | | Х | |
| Biochemistry <sup>o</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | | | Х | |
| Urinalysis <sup>p</sup> | Х | | | | | Х | | | | | | |
| INR/aPTT | Х | As | clinically in | Х | | | | | | | | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Χq | | | Χq | Х | Х |
| PK/PD Samples (see<br>Appendix 2) <sup>r</sup> | | Xr | | | Xr | | | | | | | |
| Assessment of Patient<br>Hospitalizations and/or Hospital<br>Visits | | Х | | | Х | | | Х | | | х | |
| Administration of Trastuzumab Emtansine | | D 2 <sup>s</sup> | | | D 1s | | | D 1s | | | | |
| Administration of Capecitabine | | D 1 | х | | | <b>–14</b> | | D 1 | <b>–14</b> | | | |
| Overall Survival | × | | X X X X X X D 2 <sup>s</sup> D 1 <sup>s</sup> D 1-14 D 1-14 | | | | | | | Х | Х | |
| Randomization into the Phase II Part of the Study | X <sup>t</sup> | | | | | | | | | | | |

# Study MO28230

# Appendix 1 Schedule of Assessments (cont.)

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

- 1. NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within **14 days** prior to first treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1).
- 2. All patients will be followed-up every 6 months (except for pregnancy, which is at 3 and 6 months after safety follow-up visit until disease progresses for tumor assessment or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than disease progression PD will continue to undergo tumor assessments every 3–6 months.
- a) Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests.
- b) HER2-positivity is defined as IHC 3+ or gene amplification by ISH. It will be performed locally for patients with mBC.
- c)Limited symptom-directed physical examination.
- d) Height to be obtained at screening or at Cycle 1 Day 1 only.
- e) Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f) Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to first study treatment.
- g) During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h) Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatment-related AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i) Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, between Days 15 and 21 in cycles 1 and 3, and between Days 15 and 21 and on Days 15 21 of Cycle 1, Cycle 3, 30 42 and on day 21 of every third cycle thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

# Appendix 1 Schedule of Assessments (cont.)

- j) Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than PD, continued tumor assessments according to the protocol every 3–6 months until PD, withdrawal of consent, or study terminaton (whichever occurs earlier).
- k)Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 4 months) as detailed in Section 4.5.1.4 of the protocol and in Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- I) An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- m) Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and white blood cells (WBC) with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils.
- n) Assessments should be performed at screening, on Day 1, 8 and 15 of Cycles 1–3, on Day 1 of all subsequent cycles, and weekly following any hematologic AE. If capecitabine is discontinued due to toxicity, assessments should be performed weekly (minimum) until resolution of the AE (Grade ≤ 1/ baseline), and on Day 1 of subsequent cycles thereafter. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- o) Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, blood urea nitrogen (BUN)/urea (mandatory), creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN).
- p) Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.

Study MO28230

# Appendix 1 Schedule of Assessments (cont.)

- q) Serum β-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.
- r) Pharmacokinetic assessments will be performed during the Dose-MTD-Finding part of the study only (see Appendix 2).
- s)Trastuzumab emtansine will be administered on Day 1 of each 3-weekly cycle for all patients with mBC in Cohort 1 and Randomized Phase II period of the study except in the first cycle where trastuzumab emtansine will be given on Day 2 (to allow PK sampling).
- t) Patients will be randomized only in the Randomized Phase II part of the study. No blinding will be used, as this is an open-label study. A 2:1 randomization ratio will be applied to allow more patients to be exposed to the combination of T DM1 and capecitabine, and to enable a more thorough assessment of the corresponding safety profile.

# Appendix 1 Schedule of Assessments (cont.)

# Table 2 Schedule of assessments for patients with LA/mGC (Phase I, Cohort 2)

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | Сус | le 4 Onw | ards | Safety<br>Follow-Up<br>Visit | Follow-<br>Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28–42 days<br>after last<br>dose | every 3–6<br>months |
| Informed Consent | Xa | | | | | | | | | | | |
| HER2 Status | Xp | | | | | | | | | | | |
| Medical History and<br>Demographics | Х | | | | | | | | | | | |
| Complete Physical Examination | Х | | | | | | | | | | | |
| Limited Physical Examination <sup>c</sup> | | Х | | | Х | | | Х | | | Х | |
| Height and Weight <sup>d</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Vital Signs <sup>e</sup> | Х | Х | | | Х | | | Х | | | Х | |
| ECOG Performance Status | Х | Х | | | Х | | | Х | | | Х | |
| Concomitant Medication Reporting | Xf | Х | | | | | Ongoi | ng | | | | |
| AE Reporting | Χg | | | | | Ongoing | | | | | Х | X <sup>h</sup> |
| 12-lead ECG | Х | | | | | | | | | | | |
| ECHO/MUGA <sup>i</sup> | Xi | | | Xi | | | Xi | | | Xi | Xi | |
| Tumor Assessments <sup>j</sup> | Х | | | | | | | | s of dose<br>occurs ea | | х | |
| Brain CT or MRIk | Х | | At th | ne discreti | on of the | investigat | or, if clinic | cally indica | ated, until | <del>disease p</del> | progression PD | |

| Bone Scan/Imaging <sup>l</sup> | Х | | | | | | As clinicall | y indicate | ed | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Hematology <sup>m</sup> | Х | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | Xn | Xn | Xn | Xn | Xn | Xn | Х | |
| Biochemistry <sup>o</sup> | Х | Xn | Xn | Xn | Xn | Xn | Xn | Xn | Xn | Xn | Х | |
| Urinalysis <sup>p</sup> | Х | | | Х | | | | | | | | |
| INR/aPTT | Х | As | As clinically indicated As clinically indicated, e.g. for patients receiving anticoagulation therapy | | | | | | | | | |
| Pregnancy Test <sup>q</sup> | Х | | | | | | Xq | | | Xq | Х | Х |
| PK/PD Samples (see<br>Appendix 2) | | x | | | Х | | | | | | | |
| Assessment of Patient<br>Hospitalizations and/or<br>Hospital Visits | | х | | | х | | | Х | | | х | |
| Administration of Trastuzumab Emtansine | | D 2 <sup>r</sup> | Х | х | Х | х | х | х | Х | х | | |
| Administration of Capecitabine | | D 1- | -14 | | D 1 | -14 | | D 1 | -14 | | | |
| Overall Survival | X | | | | | Х | | | | | Х | Х |

AE = Adverse Event; aPTT = Activated Partial Thromboplastin Time; CT = Computed Tomography; ECHO = Echocardiogram; ECOG = Eastern Cooperative Oncology Group; D= Day; INR = International Normalized Ratio; MRI = Magnetic Resonance Imaging; MUGA = Multiple-Gated Acquisition; PD = Progressive Disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; SAE = Serious Adverse Event

# Kadcyla (RO5304020) Roche Clinical Study Report - Protocol MO28230

# Appendix 1 Schedule of Assessments (cont.)

- 1. NOTE: Local laboratory (hematology, biochemistry, urinalysis, INR and aPTT assessments) at Screening: to be performed within **14 days** prior to first study treatment. Screening laboratory assessments may be done on the same day of first study treatment (Cycle1 Day1) visit.
- 2. All patients will be followed-up every 6 months (except for pregnancy, which is at 3 and 6 months after safety follow-up visit) until disease progresses for tumor assessment or study closure, whichever occurs first. Patients who discontinue study treatment for reasons other than disease progressionPD will continue to undergo tumor assessments every 3–6 months.
- a) Informed consent may be obtained at any time (including prior to the 28-day screening period) but must be obtained prior to the performance of any screening assessments. Results of screening tests or examinations performed as standard of care prior to obtaining informed consent and within 28 days prior to first study treatment may be used rather than repeating required tests.
- b) HER2-positivity is defined as IHC 3+ alone or IHC 2+ in combination with gene amplification by ISH. For patients with mGC enrolled into Cohort 2, central confirmation of HER2 status is required.
- c)Limited symptom-directed physical examination.
- d) Height to be obtained at screening or at Cycle 1 Day 1 only.
- e) Vital signs should be obtained and reviewed but are not required to be entered into the eCRF. Abnormal vital signs at any time during the course of study treatment should be recorded as AEs or SAEs.
- f) Record all prior investigational, anti-cancer therapies and concomitant medications within 28 days prior to fist study treatment.
- g) During screening, only SAEs considered related to protocol-mandated procedures will be collected.
- h) Patients will be followed for new or worsening AEs for 28 days following the last infusion of study drug or until the early termination visit, until treatment-related AEs resolve or stabilize, or until the initiation of another anti-cancer therapy, whichever occurs first. After 28 days following last study treatment administration, the investigator should continue to follow all unresolved study-related AEs and SAEs until their resolution or stabilization, the patient is lost to follow-up or until it is determined that the study treatment or participation is not the cause of the AE/SAE. Additionally, patients will be contacted regarding the occurrence of any new SAE considered to be treatment-related at 60 and 90 days following the last study treatment administration or until initiation of another anti-cancer therapy, whichever occurs first.
- i) Cardiac monitoring (ECHO/MUGA) will be performed in all patients enrolled in the study. Assessments will occur during the screening period, between Days 15 and 21 in cycles 1 and 3, and between Days 15 and 21 and on Days 15. 21, 30. 42 and 9 weeks of every 3rd cycle thereafter. ECHO or MUGA will be performed following study treatment discontinuation only if the most recent follow-up ECHO/MUGA was performed ≥ 28 days after last study treatment administration or if no post-treatment evaluation was performed.

i)

# Appendix 1 Schedule of Assessments (cont.)

- k)Tumor assessments (± 5 business days), including a CT or MRI with contrast of the chest, abdomen, and pelvis should be performed according to the indicated schedule. Tumor assessments obtained within 28 days prior to first study treatment may be used for screening purposes. Tumor response must be assessed through physical examination and imaged-based evaluation using RECIST version 1.1. Assessments should include an evaluation of all sites of disease. In cases where there is suspicion of progression before the next scheduled assessment, an unscheduled assessment should be performed. The same radiographic procedure used to define measurable disease sites at baseline must be used throughout the study, e.g. the same contrast protocol for CT scans. For patients who discontinue study treatment for reasons other than PD, continued tumor assessments according to the protocol every 3–6 months until PD, withdrawal of consent, or study termination (whichever occurs earliest).
- I) Patients with isolated brain metastases may continue study treatment if they demonstrate clinical benefit (CR or PR of any duration or SD ≥ 4 months) as detailed in Section 4.5.1.4 of the protocol and in Appendix 3. A brain MRI or CT should be performed along with regularly scheduled tumor assessments in these instances.
- m) An isotope bone scan and/or other radiographic modalities (as a consequence of the anticipated Tc-99 shortage), will be performed at screening and should be repeated in the event of clinical suspicion of progression of existing bone lesions and/or the development of new bone lesions. If an isotope-based scan was performed > 28 days but ≤ 60 days prior to first study treatment, non-isotopic radiographic modalities should be utilized to document the extent of bony metastatic disease. Refer to Appendix 4 in the protocol for additional details.
- n) Hematologic assessments include Hemoglobin (Hb), hematocrit, red blood cell count, platelet count, and WBC with differential (including neutrophils, lymphocytes, monocytes, eosinophils and basophils).
- o) Assessments should be performed at screening, on Day 1, 8 and 15 of all cycles. All assessments should be performed within 72 hours preceding administration of study treatment; results must be reviewed and documented prior to administration of study treatment.
- p) Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, BUN/urea (mandatory), creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN).
- q) Includes specific gravity, pH, protein, glucose, blood, ketones and bilirubin.
- r) Serum b-HCG test must be performed during screening. Urine β-HCG test must be performed at subsequent time points for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for women not meeting the definition of postmenopausal. Testing should be performed at a local laboratory within 7 days prior to the first administration of study medication (Cycle 1, Day1). For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential. Urine pregnancy test in women of childbearing potential every
- 3 cycles and at 3 and 6 months after the safety follow-up visit. All positive urine pregnancy tests must be confirmed by a serum β-HCG test.

s)Trastuzumab emtansine will be administered on Day 1 of each weekly cycle for all patients enrolled in Cohort 2 (A&B) except in the first cycle where trastuzumab emtansine will be given on DAY 2 (to allow drug interaction assessment).

#### **PROTOCOL**

TITLE: PHASE I STUDY OF THE COMBINATION OF

TRASTUZUMAB EMTANSINE (T-DM1) AND

CAPECITABINE IN HER2-POSITIVE METASTATIC BREAST CANCER AND HER2-POSITIVE LOCALLY ADVANCED/METASTATIC GASTRIC CANCER PATIENTS, FOLLOWED BY A RANDOMIZED,

**OPEN-LABEL PHASE II STUDY OF** 

TRASTUZUMAB EMTANSINE AND CAPECITABINE VERSUS TRASTUZUMAB EMTANSINE ALONE IN HER2-POSITIVE METASTATIC BREAST CANCER

PROTOCOL NUMBER: MO28230

**EUDRACT NUMBER:** 2012-001547-46


Capecitabine (RO091978)

MEDICAL MONITOR: MD

**SPONSOR:** F. Hoffmann-La Roche Ltd

**DATE FINAL:** Version: 30-Jun-2014

**DATE AMENDED:** Version: 23-Mar-2016

# PROTOCOL AMENDMENT APPROVAL


The information contained in this document, especially any unpublished data, is the property of F. Hoffmann-La Roche Ltd (or under its control) and therefore is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Ethics Committee or Institutional Review Board. It is understood that this information will not be disclosed to others without written authorization from Roche except to the extent necessary to obtain informed consent from persons to whom the drug may be administered.

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd Protocol MO2823<mark>0</mark>4, Version 4

# PROTOCOL AMENDMENT, VERSION 4 RATIONALE

Changes to the protocol have been made according to the latest clinical information and current recommendations. Specifically, the section on risks associated with capecitabine has been updated following the inclusion of the contraindication in the capecitabine SmPC for patients with known complete absence of dihydropyrimidine dehydrogenase (DPD) activity, and to include additional side effects (ophthalmological complications, acute renal failure from dehydration) and the risk of leucovorin which may increase the toxicity of capecitabine. The safety reporting of pregnancies has also been updated to highlight information that will be requested by Roche Drug Safety.

The sections on Assessment of causality of new adverse events, Adverse events occurring secondary to other events, Deaths and Pre-existing medical conditions have been updated according to the latest Roche guidance, and new sections describing the reporting of Abnormal vital sign values, Abnormal liver function tests, and Adverse events associated with an overdose or error in drug administration have been added.

The medical monitor and statistician for the study have been replaced.

The number of patients in the Randomized Phase II study has been reduced, due to slow recruitment and difficulty finding patients.

Minor changes have been made to inclusion criterion (to improve clarity and to align the synopsis and protocol), exclusion criterion (to reflect changes in treatment practice following the regulatory approval of trastuzumab emtansine).

As vital signs are not recorded in the eCRF, there are no data to summarize and so this information has been deleted from the statistical analyses.

Deleted text appears in <del>black strikethrough</del>. New text is marked with <del>yellow highlighting</del>. This amendment represents cumulative changes to the original protocol.

# PROTOCOL AMENDMENT, VERSION 4 SUMMARY OF CHANGES

| PROTOCOL Title Page | | |
|-------------------------|----|-----|
| MEDICAL MONITOR: | MD | -MD |
| FINAL PROTOCOL APPROVAL | | |

# **SYNOPSIS**

# Study Design

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

Approximately 160 210 additional patients with HER2-positive mBC will be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to the Phase II part of the study; however, they will be followed up until end of study (EOS).

# **Duration of treatment and follow-up**

All patients will be treated until investigator-assessed disease progression, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor. In case of toxicities requiring the discontinuation of capecitabine, single agent trastuzumab emtansine may be continued. In case of toxicities requiring the discontinuation of trastuzumab emtansine, the patient will be followed up until EOS (treatment with capecitabine alone is not allowed). If toxicity is considered by the investigator to be related to only one of the two agents, the non implicated agent can be continued as single-agent therapy.

#### **Number of Patients**

Randomized Phase II: Exploration of Efficacy and Safety in mBC Exploration of efficacy and safety in mBC will be based on approximately 160 210 randomized patients in total.

#### Inclusion Criteria

#### For mBC Patients

17. Disease progression on at least one prior regimen containing trastuzumab and chemotherapy either separately or in combination. Patients may be eligible to receive study therapy in the first-line setting if trastuzumab and chemotherapy were given in the [neo]adjuvant setting.

# **Exclusion Criteria**

#### For mBC Patients

- 2. Prior treatment with trastuzumab emtansine or prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine.
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogues, such as brivudine
  - b) Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
  - Known complete absence of dihyropyrimidine dehydrogenase (DPD) activity. Signs or symptoms suggesting that the patient has dihydropyrimidine dehydrogenase (DPD) deficiency

#### For LA/mGC Patients

- 2. Prior treatment with trastuzumab emtansine or prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine.
- 5. Related capecitabine contraindications:
  - a) Treatment with sorivudine or its chemically-related analogues, such as brivudine
  - b) Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
  - c) Known complete absence of DPD activity. Signs or symptoms suggesting that the patient has DPD deficiency

# **Safety Outcome Measures**

Vital signs and ECOG performance status

#### **Safety Endpoints:**

# Phase I, Cohort 1: MTD-Finding: mBC

LVEF over time will be summarized as mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

# Randomized Phase II: Exploration of Safety in mBC

Safety endpoints during the Randomized Phase II part of the study will be assessed via: total AEs, Grade ≥ 3 AEs, SAEs, premature withdrawal from study medication, AESIs, events to monitor, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

# Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd

Protocol MO28230, Version 4

LVEF over time will be summarized as mean, median and range (minimum and maximum) and will be presented graphically. Vital signs will be analyzed in a similar way.

# **Determination of Sample Size**

# Sample Size for Randomized Phase II: Exploration of Efficacy and Safety in mBC

The sample size for the primary endpoint BOR is based on a Fisher's exact test with an alpha level of 5% (one-sided), power of 70% 80% and the clinical assumption of a BOR rate of 43% with trastuzumab emtansine alone and 62.5% with the combination of trastuzumab emtansine and capecitabine. Approximately 160 210 patients (approximately 80 105 patients in each treatment group), including a 15% withdrawal rate, will be randomized with a 1:1 ratio to either trastuzumab emtansine alone or the combination of trastuzumab emtansine and capecitabine.

# **SECTION 3: STUDY DESIGN**

## 3.1.1 OVERVIEW OF STUDY DESIGN

{...}

# **Duration of Treatment and Patient Follow-up**

<u>Duration of treatment:</u> All patients will be treated until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor. In case of toxicities requiring the discontinuation of capecitabine, single agent trastuzumab emtansine may be continued. In case of toxicities requiring the discontinuation of trastuzumab emtansine, the patient will be followed up until EOS (treatment with capecitabine alone is not allowed). If toxicity is considered by the investigator to be related to only one of the two agents, the non-implicated agent can be continued as single agent therapy.

# **Duration of Study, Database Closure and Data Reporting**

{...}

Figure 1 Overview of Study Design



<sup>&</sup>lt;sup>1</sup> Capecitabine doses are administered daily on Days 1–14 q3w

mBC = metastatic breast cancer; LA/mGC = locally advanced/metastatic gastric cancer; MTD = maximum tolerated dose; q3w = every 3 weeks; qw = weekly.

# 3.1.1.2 Overview of Phase II: Exploration of Efficacy and Safety in Patients with mBC

{...}

Approximately 160 210 additional patients with HER2-positive mBC will be randomized into the Phase II part of the study. Patients in the Phase I part of the study will not contribute to the Phase II part of the study; however, they will be followed-up until end of study (EOS).

# 3.1.1.4 Number of Patients

Overall, it is anticipated that the maximum number of patients enrolled into the study will be approximately 190 240.

**Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd** Protocol MO28230, Version 4

6

<sup>&</sup>lt;sup>2</sup> The MTD defined in the mBC Phase I study will be implemented in the mBC Randomized Phase II and mGC Phase I studies

<sup>&</sup>lt;sup>3</sup> Cohort 2 will open to recruit patients with LA/mGC using the MTD defined in Phase I for patients with mBC. Dose Level 1 will not be explored in Cohort 2 (see also Section 3.3.2.2)

<sup>&</sup>lt;sup>4</sup> Stratification factor: Number of prior lines of treatment for metastatic disease (≤1 or >1; excluding single-agent hormones)

{...}

# Randomized Phase II: Exploration of Efficacy and Safety in mBC

For this part of the study, a total of approximately 160 210 patients with mBC will be randomized.

{...}

# 3.4.2.4 Secondary Safety Outcome Measures

{...}

• Vital signs and ECOG performance status

{...}

# 3.4.3.3 Secondary Safety Outcome Measures

{...}

• Vital signs and ECOG performance status

{...}

## **SECTION 4: MATERIALS AND METHODS**

#### 4.1.3 INCLUSION CRITERIA

#### 4.1.3.1 For Patients with mBC

Patients must meet the following criteria for study entry:

{...}

17. Disease progression on at least one prior regimen containing trastuzumab and chemotherapy either separately or in combination. Patients may be eligible to receive study therapy in the first-line setting if trastuzumab and chemotherapy were given in the [neo]adjuvant setting.

{...}

#### 4.1.3.2 For Patients with LA/mGC

Patients must meet the following criteria for study entry:

{...}

12. Life expectancy ≥12 weeks

{...}

# Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd Protocol MO28230, Version 4

# 4.1.4 EXCLUSION CRITERIA

#### 4.1.4.1 For Patients with mBC

{...}

2. Prior treatment with trastuzumab emtansine or prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine

{...}

- 5. Related capecitabine contraindications:
- a) Treatment with sorivudine or its chemically-related analogues, such as brivudine
- b) Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
- c) Known complete absence of DPD activity. Signs or symptoms suggesting that the patient has DPD deficiency

{...}

#### 4.1.4.2 For Patients with LA/mGC

{...}

2. Prior treatment with trastuzumab emtansine or prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine

{...}

- 5. Related capecitabine contraindications:
- a) Treatment with sorivudine or its chemically-related analogues, such as brivudine
- b) Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
- c) Known complete absence of DPD activity. Signs or symptoms suggesting that the patient has DPD deficiency

# **SECTION 5: ASSESSMENT OF SAFETY**

# 5.1.2 RISKS ASSOCIATED WITH CAPECITABINE

{...}

RarelyA rare, unexpected, severe toxicity (e.g. stomatitis, diarrhea, mucosal inflammation, neutropenia, and neurotoxicity) associated with 5-FU has been attributed to deficiency of dihydropyrimidine dehydrogenase (DPD) activity. Therefore, a link between decreased levels of DPD and increased, potentially fatal, toxic effects of 5-FU cannot be excluded. Patients with low or absent DPD activity, an enzyme involved in fluorouracil degradation, are at increased risk for severe, life-threatening, or fatal adverse reactions caused by fluorouracil.

Although DPD deficiency cannot be precisely defined, it is known that patients with certain homozygous or certain compound heterozygous mutations in the *DPYD* gene locus, which can cause complete or near complete absence of DPD enzymatic activity (as determined by laboratory assays), have the highest risk of life-threatening or fatal toxicity<sup>47</sup> and should not be treated with capecitabine. No dose has been proven safe for patients with complete absence of DPD activity.

For patients with partial DPD deficiency (such as those with heterozygous mutations in the *DPYD* gene) and where the benefits of capecitabine are considered to outweigh the risks (taking into account the suitability of an alternative non-fluoropyrimidine chemotherapeutic regimen), these patients must be treated with extreme caution, and frequent subsequent monitoring and dose adjustment according to toxicity. There is insufficient data to recommend a specific dose in patients with partial DPD activity as measured by specific test.

In patients with unrecognized DPD deficiency treated with capecitabine, life-threatening toxicities manifesting as acute overdose may occur. In the event of Grade 2–4 acute toxicity, treatment must be discontinued immediately. Permanent discontinuation should be considered based on clinical assessment of the onset, duration, and severity of the observed toxicities.

Capecitabine can induce hand-foot syndrome (palmar-plantar erythrodysesthesia or chemotherapy-induced acral erythema), which is a cutaneous toxicity. Persistent or severe hand-foot syndrome (Grade 2 and above) can eventually lead to loss of fingerprints, which could impact patient identification. For patients receiving capecitabine monotherapy in the metastatic setting, the median time to onset was 79 days (range 11–360 days), with a severity range of Grades 1 to 3. Grade 1 hand-foot syndrome is defined by numbness, dysesthesia/paresthesia, tingling or erythema of the hands and/or feet and/or discomfort which does not disrupt normal activities. Grade 2 is defined as painful erythema and swelling of the hands and/or feet and/or discomfort affecting the patient's activities of daily living (ADL). Grade 3 is defined as moist desquamation, ulceration, blistering or severe pain of the hands and/or feet and/or severe discomfort that causes the patient to be unable to work or perform

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd Protocol MO28230, Version 4

ADL. If Grade 2 or 3 hand-foot syndrome occurs, administration of capecitabine should be interrupted until the event resolves or decreases in intensity to Grade 1. Following Grade 3 hand-foot syndrome, subsequent doses of capecitabine should be decreased.

Patients should be carefully monitored for ophthalmological complications such as keratitis and corneal disorders, especially if they have a prior history of eye disorders. Treatment of eye disorders should be initiated as clinically appropriate.

Capecitabine can induce hyperbilirubinemia. Administration of capecitabine should be interrupted if treatment-related elevations in bilirubin of  $> 3.0 \times ULN$  or treatment-related elevations in hepatic aminotransferases (ALT/AST) of Grade  $\geq 2$  occur.

Dehydration may cause acute renal failure, especially in patients with preexisting compromised renal function or when capecitabine is given concomitantly with known nephrotoxic agents. Acute renal failure secondary to dehydration might be potentially fatal.

Capecitabine can induce severe skin reactions such as Stevens-Johnson syndrome and toxic epidermal necrolysis. Capecitabine should be permanently discontinued in patients who experience a severe skin reaction possibly attributable to capecitabine during treatment.

Leucovorin affects the pharmacodynamics of capecitabine and may increase the toxicity of capecitabine. This may be relevant in patients receiving folic acid supplementation for folate deficiency due to the similarity between folinic acid and folic acid.

# 5.1.4 DEFINITION OF DOSE-LIMITING TOXICITY

{...}

# Non-hematologic

{...}

8. Grade 2 toxicity requiring interruption of treatment for > 14 days

NOTE: Patients experiencing acute early-onset (within 1 week) or unusually severe toxicity of Grade ≥ 3 hand-foot syndrome, diarrhea, mucositisstomatitis, mucosal inflammation, neurotoxicity, neutropenia, or febrile neutropenia with ANC < 500 cells/mm³ during Cycle 1 must be tested for DPD deficiency (a central laboratory will be appointed). The SC will adjudicate in cases of DLTs that are not covered by the existing DLT criteria.

# 5.3.4 ASSESSMENT OF CAUSALITY OF ADVERSE EVENTS

Investigators should use their knowledge of the patient, the circumstances surrounding the event, temporal relationship of event onset to the initiation of study drug, course of the event considering especially the effects of dose reduction or discontinuation of study drug or reintroduction of study drug (as applicable), known association of the event with the study drug or with similar treatments, known association of the event with the disease under study, presence of risk factors in the patient or use of concomitant medications known to increase the occurrence of the event, presence of non-treatment-related factors that are known to be associated with the occurrence of the event, and an evaluation of any potential alternative causes to determine whether or not an AE is considered to be related to study drugs, indicating "yes" or "no" accordingly.

{...}

# 5.3.5 PROCEDURES FOR RECORDING ADVERSE EVENTS

# 5.3.5.2 Adverse Events Occurring Secondary to Other Events

{...}

However, medically significant AEs occurring secondary to an initiating event that are separated in time should be recorded as independent events on the eCRF. For example, if a severe gastrointestinal hemorrhage leads to renal failure, both events should be recorded separately on the eCRF. All AEs should be recorded separately on the Adverse Event eCRF if it is unclear whether the events are associated.

# 5.3.5.5 Abnormal Vital Sign Values

Not every vital sign abnormality qualifies as an AE. A vital sign result must be reported as an AE if it meets any of the following criteria:

- Is accompanied by clinical symptoms
- Results in a change in study treatment (e.g., dosage modification, treatment interruption, or treatment discontinuation)
- Results in a medical intervention or a change in concomitant therapy
- Is clinically significant in the investigator's judgment

It is the investigator's responsibility to review all vital sign findings. Medical and scientific judgment should be exercised in deciding whether an isolated vital sign abnormality should be classified as an AE.

If a clinically significant vital sign abnormality is a sign of a disease or syndrome (e.g., high blood pressure), only the diagnosis (i.e., hypertension) should be recorded on the Adverse Event eCRF.

Observations of the same clinically significant vital sign abnormality from visit to visit should only be recorded once on the Adverse Event eCRF (see Section 5.3.5.3 for details on recording persistent AEs).

# 5.3.5.6 Abnormal Liver Function Tests

The finding of an elevated ALT or AST ( $>3 \times$  baseline value) in combination with either an elevated total bilirubin ( $>2 \times$  ULN) or clinical jaundice in the absence of cholestasis or other causes of hyperbilirubinemia is considered to be an indicator of severe liver injury (as defined by Hy's law). Therefore, investigators must report as an AE the occurrence of either of the following:

- Treatment-emergent ALT or AST > 3 × baseline value in combination with total bilirubin > 2 × ULN (of which ≥ 35% is direct bilirubin)
- Treatment-emergent ALT or AST > 3 × baseline value in combination with clinical jaundice

The most appropriate diagnosis or (if a diagnosis cannot be established) the abnormal laboratory values should be recorded on the Adverse Event eCRF (see Section 5.3.5.4) and reported to the Sponsor immediately (i.e., no more than 24 hours after learning of the event), either as an SAE or a non-serious AE of special interest (see Section 5.4.2).

#### 5.3.5.7 Deaths

{...}

Death should be considered an **outcome** and not a distinct event. The event or condition that caused or contributed to the fatal outcome should be recorded as the single medical concept on the AE eCRF. Generally, only one such event should be reported. If the cause of death is unknown and cannot be ascertained at the time of reporting, "**unexplained death**" should be recorded on the AE eCRF. If the cause of death later becomes available (e.g., after autopsy), "unexplained death" should be replaced by the established cause of death. The term "**sudden death**" should be used only for the occurrence of an abrupt and unexpected death due to presumed cardiac causes in a patient with or without preexisting heart disease, within 1 hour after the onset of acute symptoms or, in the case of an unwitnessed death, within 24 hours after the patient was last seen alive and stable.

{...}

# 5.3.5.8 Pre-Existing Medical Conditions

A pre-existing medical condition is one that is present at the start of this study. Such conditions should be recorded on the Medical and Surgical History eCRF.

A pre-existing medical condition should be recorded as an AE <u>only</u> if the frequency, severity, or character of the condition worsens during the study. When recording such events on the AE eCRF, it is important to convey the concept that

Trastuzumab Emtansine-F. Hoffmann-La Roche Ltd Protocol MO28230, Version 4

the pre-existing condition has changed by including applicable descriptors (e.g., "more frequent headaches" or "worsening gastrointestinal reflux disease").

# 5.3.5.11 Adverse Events Associated with an Overdose or Error in Drug Administration

An overdose is the accidental or intentional use of a drug in an amount higher than the dose being studied. An overdose or incorrect administration of study treatment is not itself an AE, but it may result in an AE. All overdose or incorrect administrations of study drug with/without AEs associated should be recorded on the AE eCRF. If the associated AE fulfills seriousness criteria, the event should be reported to the Sponsor immediately (i.e., no more than 24 hours after learning of the event; see Section 5.4.2).

# 5.4.3 REPORTING REQUIREMENTS FOR PREGNANCIES

# **5.4.3.1** Pregnancies in Female Patients

{...}

Additional information on any trastuzumab emtansine-exposed pregnancy and infant will be requested by Roche Drug Safety at specific time points (i.e., after having received the initial report, at the end of the second trimester, 2 weeks after the expected date of delivery, and at 3, 6, and 12 months of the infant's life).

Any serious adverse events associated with the pregnancy (e.g., an event in the fetus, an event in the mother during or after the pregnancy, or a congenital anomaly/birth defect in the child) should be reported on the Adverse Event eCRF. In addition, the investigator will submit a Clinical Trial Pregnancy Reporting Form when updated information on the course and outcome of the pregnancy becomes available.

# 6.1 DETERMINATION OF SAMPLE SIZE

# Sample Size for Randomized Phase II: Exploration of Efficacy and Safety in mBC

The sample size for the primary endpoint BOR is based on a Fisher's exact test with an alpha level of 5% (one-sided), 48,4950,51 power of 70% 80% and the clinical assumption of a BOR rate of 43% with trastuzumab emtansine alone and 62.5% with the combination of trastuzumab emtansine and capecitabine. Approximately 160 210-patients (approximately 80 105 patients in each treatment group), including a 15% withdrawal rate, will be randomized with a 1:1 ratio to trastuzumab emtansine alone or the combination of trastuzumab emtansine and capecitabine.

# 6.5 SAFETY ANALYSES

# Safety Population Phase I, Cohort 1: mBC

{...}

LVEF will be summarized over time using mean, median and range (minimum and maximum) and will be presented graphically. <del>Vital signs will be analyzed in a similar way.</del>

{...}

# Randomized Phase II: Exploration of Safety in mBC

{...}

Safety endpoints during Phase II will be assessed via total AEs, Grade ≥3 AEs, SAEs, AESIs (as described in Section 5), fatal AEs and their causes, events to monitor, premature withdrawal from study medication and/or study, laboratory parameters, LVEF, exposure to study medication, concomitant medications, vital signs, ECOG performance status, and physical examination.

{...}

LVEF will be summarized over time using mean, median and range (minimum and maximum) and will be presented graphically. <del>Vital signs will be analyzed in a similar way.</del>

{...}

# 6.9 INTERIM ANALYSES

{...}

The IDMC will also monitor safety outcomes after 25, 75, and 150 patients have received at least 3 cycles (Cycle 3 Day 21) of treatment in the Randomized Phase II part of the study.

{...}

#### 10. REFERENCES

- 47. Amstutz U, Froehlich TK, Largiadèr CR. Dihydropyrimidine dehydrogenase gene as a major predictor of severe 5-fluorouracil toxicity. Pharmacogenomics 2011;12(9):1321–36.
- 48. Drug Safety Report Xeloda and Fingerprint loss, 1067787, January 2016 (CDS Vs 14.0).

# Appendix 1 Schedule of Assessments

# Table 1 Schedule of assessments for mBC patients (Phase I, Cohort 1 and Randomized Phase II)

{...}

| | Screening <sup>1</sup> | | Cycle 1 | | | Cycle 2–3 | 3 | Cycle | e 4 Onwa | ards | Safety<br>Follow-Up<br>Visit | Follow-<br>Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 3-6<br>months |
| Administration of Capecitabinet | | D 1 | D 1–14 | | D 1–14 | | | D 1–14 | | | | |
| Randomization into the Phase II Part of the Study | X <mark>ŧu</mark> | | | | | | | | | | | |

{...}

- o) Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, blood urea nitrogen (BUN)/urea (mandatory), creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN). Fasting is required before biochemistry assessment.
- t) Capecitabine must be given within 30 minutes after a meal.

# Trastuzumab Emtansine

# **Appendix 1** Schedule of Assessments (cont.)

# Table 2 Schedule of assessments for patients with LA/mGC (Phase I, Cohort 2)

{...}

| | Screening <sup>1</sup> | | Cycle 1 | | ( | Cycle 2–3 | 3 | Cycle | e 4 Onwa | ırds | Safety<br>Follow-Up<br>Visit | Follow-<br>Up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 1 | 8 | 15 | 1 | 8 | 15 | 28-42 days<br>after last<br>dose | every 3-6<br>months |
| Administration of Capecitabines | | D 1 | D 1–14 | | D 1–14 | | | D 1–14 | | | | |

- o) Biochemistry assessments include: sodium, potassium, chloride, calcium, magnesium, glucose, blood urea nitrogen (BUN)/urea (mandatory), creatinine, uric acid, total protein, albumin, alkaline phosphatase, ALT (SGPT), AST (SGOT), G-GT, LDH, total bilirubin (and direct bilirubin where total bilirubin > ULN). Fasting is required before biochemistry assessment.
- s) Capecitabine must be given within 30 minutes after a meal.